CLINICAL TRIAL: NCT04403880
Title: Characterizing SARS-CoV-2-specific Immunity in Convalescent Individuals
Brief Title: Characterizing SARS-CoV-2-specific Immunity in Individuals Who Have Recovered From COVID-19
Status: Completed | Type: Observational
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Other Study IDs: HVTN 405/HPTN 1901; 5UM1AI068614-14 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Persons not hospitalized for COVID-19, without clinical spectrum or outcomes specified in group 3
  * 1A: Persons with asymptomatic infection, ages 18 through 55, inclusive
  * 1B: Persons with asymptomatic infection, age > 55
  * 1C: Persons with symptomatic infection (ie, COVID-19) ages 18 through 55
  * 1D: Persons with symptomatic infection (ie, COVID-19), age > 55
  Interventions: Other: Sample collection
- Group 2: Persons previously hospitalized for COVID-19, without clinical spectrum or outcomes specified in group 3
  * 2A: Persons 18 through 55 years of age
  * 2B: Persons > 55 years of age
  Interventions: Other: Sample collection
- Group 3: Persons with specific clinical spectrums or outcomes, regardless of hospitalization history (eg, persons recovered after intubation, with prolonged viral shedding, with myocarditis/pericarditis, with rapid recovery from COVID-19, with a second positive SARS-CoV-2 RT-PCR test result after a negative result)
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — * Optional nasal specimen(s)
  * Blood collection

SUMMARY:
The purpose of this study is to learn more about infection with and recovery from the virus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Some people know this virus by the name "coronavirus." It can cause the disease called COVID-19.

The information gained from the study will be used to help develop better tests for SARS-CoV-2 infection and COVID-19 disease and may help in developing future vaccines and treatments by allowing researchers to determine the difference between the body's immune response to natural SARS-CoV-2 infection and immunization with a SARS-CoV-2 vaccine.

DETAILED DESCRIPTION:
This study aims to characterize the SARS-CoV-2-specific immunity in convalescent individuals.

The observational cohort study will include 3 groups, as described in the table below.

Participants will complete a minimum of one visit (1-8 weeks post resolution of COVID-19 OR 2-10 weeks post most recent positive SARS-CoV-2 test, if asymptomatic) and optional visits approximately 2 months, 4 months, and 1 year later. Participants diagnosed with SARS-CoV-2 infection at an optional follow-up visit may be contacted more frequently. Additional follow up visit(s) may be added over time in response to evolving information regarding SARS-CoV-2 infection and COVID-19.

Study visits may include physical examinations, medical history, questionnaires, pregnancy tests (for participants assigned female at birth), blood draws, optional nasal samples, and optional HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Reports having had a positive test for SARS-CoV-2.
* Reports resolution of COVID-19 within 1-8 weeks of enrollment OR, if asymptomatic infection, reports positive SARS-CoV-2 test within 2-10 weeks of enrollment. Not excluded: individuals with symptoms consistent with residual sequelae of resolved COVID-19, in the clinical judgement of the investigator.
* Access to a participating HVTN or HPTN CRS and willingness to be followed for the planned duration of the study.
* Ability and willingness to provide informed consent.
* Assessment of understanding: volunteer demonstrates understanding of this study.
* Volunteers who were assigned female sex at birth: negative urine or serum beta human chorionic gonadotropin (β-HCG) pregnancy test within 4 days of enrollment visit (ie, prior to enrollment blood draw or nasal collections). Persons who are NOT of reproductive potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records) or having reached menopause (no menses for ≥ 1 year ), are not required to undergo pregnancy testing.

Exclusion Criteria:

* Reports current COVID-19.
* Pregnant.
* Receipt of SARS-CoV-2 specific antibodies (eg, convalescent plasma or sera, monoclonal antibodies, hyperimmune globulin). Not excluded: antibody therapy without SARS-CoV-2 specificity (eg, IL-6 pathway inhibitors for COVID-19).
* SARS-CoV-2 vaccine(s) received in a prior vaccine trial.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or a volunteer's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons reporting a positive test for SARS-CoV-2 and resolution of COVID-19 within 1-8 weeks of enrollment OR, if asymptomatic infection, reporting positive SARS-CoV-2 test within 2-10 weeks of enrollment.
Sampling Method: Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Corey, Study Chair — HIV Vaccine Trials Network, Fred Hutch; Shelly Karuna, Study Chair — HIV Vaccine Trials Network, Fred Hutch
Locations (53):
- United States (21):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Bridge HIV CRS, San Francisco, California
  - George Washington University CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Adolescent & Young Adult Research at The CORE Center (AYAR at CORE), Chicago, Illinois
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health Clinical Research Site CRS, Boston, Massachusetts
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Harlem Prevention Center CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Bronx Prevention Research Center CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Malawi CRS, Lilongwe, Malawi
- Peru (5):
  - San Miguel CRS, San Miguel, Lima region
  - Asociacion Civil Selva Amazonica (ACSA) CRS, Iquitos, Maynas
  - CITBM - UNIDEC, Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS, Bellavista, Provincia Constitucional del Callao
  - Via Libra CRS, Lima
  - Barranco CRS, Lima
- South Africa (22):
  - Josha Research CRS, Bloemfontein
  - Emavundleni CRS, Cape Town
  - Groote Schuur HIV CRS, Cape Town
  - Khayelitsha CRS / (CIDRI UCT), Cape Town
  - Masiphumelele Clinical Research Site (MASI) CRS, Cape Town
  - Chatsworth CRS, Chatsworth
  - Botha's Hill CRS, Durban
  - CAPRISA eThekwini CRS, Durban
  - Vulindlela CRS, Durban
  - Isipingo CRS, Isipingo
  - Kliptown Soweto CRS, Johannesburg
  - Soweto HVTN CRS, Johannesburg
  - Aurum Institute Klerksdorp CRS, Klerksdorp
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith
  - Nelson Mandela Academic Research Unit CRS, Mthatha
  - Synexus Stanza Clinical Research Centre CRS, Pretoria
  - Rustenburg CRS, Rustenburg
  - Setshaba Research Centre CRS, Soshanguve
  - Tembisa Clinic 4 CRS, Tembisa
  - The Aurum Institute Tembisa Clinical Research Centre CRS, Tembisa
  - Tongaat CRS, Tongaat
  - Verulam CRS, Verulam
- Matero Reference Clinic CRS, Lusaka, Zambia
- Zimbabwe (3):
  - St Mary's CRS, Chitungwiza
  - Zengeza CRS, Chitungwiza
  - Seke South CRS, Harare

REFERENCES:
- [Derived] Karuna S, Gallardo-Cartagena JA, Theodore D, Hunidzarira P, Montenegro-Idrogo J, Hu J, Jones M, Kim V, De La Grecca R, Trahey M, Karg C, Takalani A, Polakowski L, Hutter J, Miner MD, Erdmann N, Goepfert P, Maboa R, Corey L, Gill K, Li SS; HVTN 405/HPTN 1901 Study Team. Post-COVID symptom profiles and duration in a global convalescent COVID-19 observational cohort: Correlations with demographics, medical history, acute COVID-19 severity and global region. J Glob Health. 2023 Jun 23;13:06020. doi: 10.7189/jogh.13.06020. PMID 37352144
- [Derived] Karuna S, Li SS, Grant S, Walsh SR, Frank I, Casapia M, Trahey M, Hyrien O, Fisher L, Miner MD, Randhawa AK, Polakowski L, Kublin JG, Corey L, Montefiori D; HVTN 405/HPTN 1901 Study Team. Neutralizing antibody responses over time in demographically and clinically diverse individuals recovered from SARS-CoV-2 infection in the United States and Peru: A cohort study. PLoS Med. 2021 Dec 6;18(12):e1003868. doi: 10.1371/journal.pmed.1003868. eCollection 2021 Dec. PMID 34871308

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1A: 1A: Asymptomatic, 18 - 55
- Group 1B: 1B: Asymptomatic, > 55
- Group 1C: 1C: Symptomatic, 18 - 55
- Group 1D: 1D: Symptomatic, > 55
- Group 2A: 2A: Hospitalized, 18 - 55
- Group 2B: 2B: Hospitalized, > 55
- Group 3: 3: Clinical spectrums
Period: Overall Study
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Started | 129 | 51 | 182 | 77 | 122 | 74 | 125
Completed | 81 | 24 | 98 | 32 | 68 | 44 | 67
Not Completed | 48 | 27 | 84 | 45 | 54 | 30 | 58
Not completed — Death | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 8 | 7 | 8 | 1 | 8
Not completed — Withdrawal by Subject | 8 | 9 | 22 | 16 | 16 | 8 | 11
Not completed — Participant Unable to Adhere to Visit Schedule | 6 | 5 | 12 | 2 | 8 | 1 | 2
Not completed — Participant Unable to Comply with Study Procedure | 7 | 1 | 7 | 9 | 8 | 8 | 19
Not completed — Pregnancy | 2 | 0 | 5 | 0 | 1 | 0 | 1
Not completed — Sponsor Decision | 2 | 0 | 14 | 1 | 1 | 0 | 2
Not completed — Other | 18 | 9 | 14 | 10 | 11 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3 | Total
Number analyzed (Participants) | 129 | 51 | 182 | 77 | 122 | 74 | 125 | 760
Age, Continuous [Median (Full Range); unit: years] | 33 [18 to 55] | 62 [56 to 82] | 35 [18 to 55] | 61 [56 to 86] | 41 [20 to 55] | 62 [56 to 83] | 43 [21 to 75] | 44 [18 to 86]
Age, Customized [Count of Participants; unit: Participants]
  18 - 25 years | 26 | 0 | 21 | 0 | 10 | 0 | 6 | 63
  26 - 35 years | 54 | 0 | 74 | 0 | 34 | 0 | 26 | 188
  36 - 45 years | 28 | 0 | 52 | 0 | 36 | 0 | 39 | 155
  46 - 55 years | 21 | 0 | 35 | 0 | 42 | 0 | 27 | 125
  56 - 65 years | 0 | 35 | 0 | 59 | 0 | 54 | 23 | 171
  66 - 75 years | 0 | 11 | 0 | 13 | 0 | 13 | 4 | 41
  Over 75 years | 0 | 5 | 0 | 5 | 0 | 7 | 0 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 21 | 129 | 42 | 70 | 33 | 54 | 408
  Male | 70 | 30 | 53 | 35 | 52 | 41 | 71 | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 19 | 28 | 28 | 30 | 27 | 52 | 212
  Not Hispanic or Latino | 101 | 32 | 153 | 49 | 92 | 47 | 73 | 547
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 8 | 1 | 5 | 0 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 83 | 17 | 87 | 20 | 68 | 27 | 27 | 329
  White | 7 | 8 | 25 | 26 | 6 | 21 | 36 | 129
  More than one race | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 6
  Unknown or Not Reported | 36 | 23 | 60 | 30 | 42 | 26 | 56 | 273
Region of Enrollment [Count of Participants; unit: Participants] — non-RSA include Malawi, Mozambique, Tanzania, Zambia, and Zimbabwe
  Participants
    United States | 25 | 18 | 28 | 26 | 24 | 25 | 51 | 197
    Peru | 25 | 16 | 25 | 25 | 25 | 25 | 50 | 191
    South Africa | 64 | 14 | 98 | 21 | 57 | 19 | 14 | 287
    Non-RSA | 15 | 3 | 31 | 5 | 16 | 5 | 10 | 85

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (BAMA IgG1) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3, overall and by region and enrollment group
Time Frame: Measured at Months 0, 2, 4
Population: The 'Overall Number of Participants Analyzed' summarized the participants number in American Population (USA and Peru only), regardless the assay availability. The 'Number Analyzed' for each antigen summarized the participants number at each time point with available assay data. The 'Number Analyzed' may be smaller than 'Overall Number of Participants Analyzed' due to assay data unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 17 | 4 | 16 | 20 | 21 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Peru | 15 | 3 | 16 | 18 | 21 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 32 | 19 | 33 | 36 | 37 | 40 | 87
  2019-nCoV S/293F-50 at Month 0-Total | 26 | 11 | 33 | 33 | 36 | 39 | 86
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 15 | 15 | 17 | 16 | 16 | 15 | 38
  2019-nCoV S/293F-50 at Month 0-USA | 11 | 8 | 17 | 15 | 15 | 14 | 37
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 18 | 36
  2019-nCoV S/293F-50 at Month 2-Peru | 21 | 2 | 19 | 16 | 20 | 18 | 36
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 34 | 12 | 36 | 41 | 36 | 37 | 76
  2019-nCoV S/293F-50 at Month 2-Total | 30 | 8 | 36 | 37 | 32 | 36 | 71
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 11 | 10 | 17 | 22 | 14 | 19 | 40
  2019-nCoV S/293F-50 at Month 2-USA | 9 | 6 | 17 | 21 | 12 | 18 | 35
  2019-nCoV S/293F-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  2019-nCoV S/293F-50 at Month 4-Peru | 22 | 2 | 17 | 13 | 18 | 16 | 19
  2019-nCoV S/293F-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 33 | 29 | 45
  2019-nCoV S/293F-50 at Month 4-Total | 29 | 3 | 27 | 25 | 29 | 27 | 43
  2019-nCoV S/293F-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 13 | 13 | 26
  2019-nCoV S/293F-50 at Month 4-USA | 7 | 1 | 10 | 12 | 11 | 11 | 24
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 DB His-50 at Month 0-Peru | 21 | 3 | 23 | 20 | 22 | 25 | 49
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 49 | 48 | 50 | 97
  SARS-CoV-2 DB His-50 at Month 0-Total | 34 | 13 | 51 | 45 | 43 | 47 | 93
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 25 | 48
  SARS-CoV-2 DB His-50 at Month 0-USA | 13 | 10 | 28 | 25 | 21 | 22 | 44
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 17 | 22 | 18 | 36
  SARS-CoV-2 DB His-50 at Month 2-Peru | 20 | 2 | 17 | 16 | 20 | 18 | 36
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 37 | 39 | 36 | 37 | 78
  SARS-CoV-2 DB His-50 at Month 2-Total | 30 | 8 | 35 | 37 | 30 | 35 | 72
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 22 | 14 | 19 | 42
  SARS-CoV-2 DB His-50 at Month 2-USA | 10 | 6 | 18 | 21 | 10 | 17 | 36
  SARS-CoV-2 DB His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 16 | 19
  SARS-CoV-2 DB His-50 at Month 4-Peru | 22 | 2 | 16 | 12 | 18 | 16 | 19
  SARS-CoV-2 DB His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 32 | 29 | 45
  SARS-CoV-2 DB His-50 at Month 4-Total | 28 | 3 | 26 | 24 | 27 | 27 | 42
  SARS-CoV-2 DB His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 DB His-50 at Month 4-USA | 6 | 1 | 10 | 12 | 9 | 11 | 23
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 21 | 3 | 23 | 20 | 22 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 49 | 47 | 50 | 97
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 34 | 14 | 51 | 45 | 41 | 48 | 91
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 25 | 48
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 13 | 11 | 28 | 25 | 19 | 23 | 42
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 18 | 19 | 22 | 18 | 34
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 20 | 2 | 16 | 16 | 20 | 18 | 34
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 35 | 11 | 35 | 41 | 36 | 36 | 75
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 29 | 8 | 31 | 37 | 30 | 34 | 70
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 12 | 9 | 17 | 22 | 14 | 18 | 41
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 9 | 6 | 15 | 21 | 10 | 16 | 36
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 13 | 18 | 16 | 17
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Peru | 20 | 2 | 17 | 10 | 16 | 16 | 17
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 26 | 30 | 28 | 40
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total | 26 | 3 | 25 | 22 | 25 | 26 | 37
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 12 | 23
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-USA | 6 | 1 | 8 | 12 | 9 | 10 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 14 | 4 | 16 | 17 | 19 | 23 | 47
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 12 | 3 | 16 | 16 | 19 | 23 | 47
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 28 | 19 | 32 | 29 | 35 | 38 | 83
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 20 | 11 | 32 | 28 | 34 | 37 | 82
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 14 | 15 | 16 | 12 | 16 | 15 | 36
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 8 | 8 | 16 | 12 | 15 | 14 | 35
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 21 | 18 | 36
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 20 | 2 | 17 | 17 | 19 | 18 | 36
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 36 | 41 | 35 | 37 | 78
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 31 | 8 | 34 | 38 | 29 | 36 | 73
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 17 | 22 | 14 | 19 | 42
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 11 | 6 | 17 | 21 | 10 | 18 | 37
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 19 | 16 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Peru | 22 | 2 | 17 | 13 | 17 | 16 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 31 | 29 | 45
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total | 29 | 3 | 27 | 25 | 27 | 27 | 43
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-USA | 7 | 1 | 10 | 12 | 10 | 11 | 24
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 22 | 4 | 25 | 22 | 22 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 19 | 3 | 24 | 20 | 20 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 46 | 22 | 52 | 45 | 46 | 50 | 97
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 31 | 13 | 51 | 43 | 40 | 47 | 92
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 27 | 23 | 24 | 25 | 48
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 12 | 10 | 27 | 23 | 20 | 22 | 43
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 19 | 22 | 18 | 36
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 20 | 2 | 18 | 17 | 20 | 18 | 36
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 38 | 41 | 36 | 37 | 77
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 31 | 8 | 36 | 38 | 30 | 35 | 71
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 22 | 14 | 19 | 41
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 11 | 6 | 18 | 21 | 10 | 17 | 35
  SARS-CoV-2 S1 C His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 16 | 19
  SARS-CoV-2 S1 C His-50 at Month 4-Peru | 22 | 2 | 16 | 12 | 18 | 16 | 19
  SARS-CoV-2 S1 C His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 32 | 29 | 45
  SARS-CoV-2 S1 C His-50 at Month 4-Total | 29 | 3 | 26 | 24 | 27 | 27 | 42
  SARS-CoV-2 S1 C His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 S1 C His-50 at Month 4-USA | 7 | 1 | 10 | 12 | 9 | 11 | 23
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 21 | 3 | 23 | 20 | 22 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 47 | 22 | 53 | 49 | 47 | 50 | 97
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 36 | 16 | 51 | 45 | 42 | 49 | 92
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 23 | 25 | 48
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 15 | 13 | 28 | 25 | 20 | 24 | 43
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 21 | 2 | 19 | 19 | 22 | 17 | 35
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 19 | 2 | 18 | 17 | 20 | 17 | 35
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 32 | 11 | 36 | 41 | 35 | 36 | 74
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 28 | 8 | 35 | 38 | 31 | 35 | 71
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 11 | 9 | 17 | 22 | 13 | 19 | 39
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 9 | 6 | 17 | 21 | 11 | 18 | 36
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 16 | 13 | 18 | 16 | 17
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Peru | 23 | 2 | 15 | 11 | 16 | 16 | 17
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 25 | 26 | 30 | 28 | 41
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total | 30 | 4 | 24 | 23 | 25 | 27 | 39
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 9 | 13 | 12 | 12 | 24
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-USA | 7 | 2 | 9 | 12 | 9 | 11 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 48
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 22 | 3 | 24 | 22 | 22 | 25 | 48
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 51 | 47 | 50 | 97
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 38 | 13 | 52 | 47 | 42 | 48 | 92
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 23 | 25 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 16 | 10 | 28 | 25 | 20 | 23 | 44
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 18 | 36
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 20 | 2 | 18 | 16 | 20 | 18 | 36
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 36 | 41 | 36 | 37 | 79
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 31 | 8 | 35 | 37 | 32 | 36 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 17 | 22 | 14 | 19 | 43
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 11 | 6 | 17 | 21 | 12 | 18 | 38
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Peru | 22 | 2 | 17 | 13 | 18 | 16 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 33 | 29 | 45
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total | 29 | 3 | 27 | 25 | 29 | 27 | 43
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 13 | 13 | 26
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-USA | 7 | 1 | 10 | 12 | 11 | 11 | 24
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 14 | 4 | 16 | 17 | 19 | 24 | 48
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 12 | 3 | 16 | 16 | 19 | 24 | 48
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 28 | 19 | 32 | 30 | 35 | 39 | 85
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 22 | 11 | 32 | 29 | 33 | 38 | 82
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 14 | 15 | 16 | 13 | 16 | 15 | 37
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 10 | 8 | 16 | 13 | 14 | 14 | 34
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 17 | 36
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 20 | 2 | 17 | 17 | 20 | 17 | 36
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 35 | 12 | 37 | 41 | 35 | 34 | 75
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 30 | 7 | 35 | 38 | 30 | 33 | 68
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 12 | 10 | 18 | 22 | 13 | 17 | 39
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 10 | 5 | 18 | 21 | 10 | 16 | 32
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Peru | 22 | 2 | 17 | 14 | 18 | 16 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 32 | 29 | 45
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total | 29 | 3 | 27 | 26 | 27 | 27 | 41
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-USA | 7 | 1 | 10 | 12 | 9 | 11 | 22

2. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (BAMA IgG1) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3, overall and by region and enrollment group
Time Frame: Measured at Months 0, 2, 4
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
MFI
  2019-nCoV S/293F-1000 at Month 0-Peru: number analyzed (Participants) | 17 | 4 | 16 | 20 | 21 | 25 | 49
  2019-nCoV S/293F-1000 at Month 0-Peru | 10735 [3712.8 to 14037.2] | 5225.2 [3182.4 to 10215.2] | 22000 [10914.1 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [15797.8 to 22000]
  2019-nCoV S/293F-1000 at Month 0-Total: number analyzed (Participants) | 32 | 19 | 33 | 36 | 37 | 40 | 87
  2019-nCoV S/293F-1000 at Month 0-Total | 7790.9 [774.4 to 11902.2] | 3413.2 [1 to 9553.6] | 13862.2 [5081 to 22000] | 22000 [8377.9 to 22000] | 22000 [16996.2 to 22000] | 22000 [22000 to 22000] | 16428.8 [5858.1 to 22000]
  2019-nCoV S/293F-1000 at Month 0-USA: number analyzed (Participants) | 15 | 15 | 17 | 16 | 16 | 15 | 38
  2019-nCoV S/293F-1000 at Month 0-USA | 958.8 [1 to 7844.4] | 3013 [1 to 9553.6] | 8418 [2056.5 to 21876.8] | 9064.2 [5341.4 to 22000] | 19159.8 [6267.3 to 22000] | 22000 [20962.2 to 22000] | 8637 [2768.2 to 14335.2]
  2019-nCoV S/293F-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 18 | 36
  2019-nCoV S/293F-1000 at Month 2-Peru | 2149 [1146 to 4407.1] | 14129.9 [10194.8 to 18064.9] | 7039 [2096.1 to 11836.4] | 14945 [8318.5 to 20964.4] | 21771.9 [9814.5 to 22000] | 22000 [20542.2 to 22000] | 17594.6 [8674.8 to 22000]
  2019-nCoV S/293F-1000 at Month 2-Total: number analyzed (Participants) | 34 | 12 | 36 | 41 | 36 | 37 | 76
  2019-nCoV S/293F-1000 at Month 2-Total | 2090.9 [955.2 to 4515.9] | 3946.9 [83.3 to 8101.2] | 6997.9 [2851.1 to 13690.4] | 12310.8 [6517 to 19928.8] | 13478.1 [5632.2 to 22000] | 22000 [12489 to 22000] | 7604.6 [2817.5 to 18727.2]
  2019-nCoV S/293F-1000 at Month 2-USA: number analyzed (Participants) | 11 | 10 | 17 | 22 | 14 | 19 | 40
  2019-nCoV S/293F-1000 at Month 2-USA | 2032.8 [229.4 to 4360.1] | 1315.8 [46.9 to 6980.1] | 5189.8 [3272.8 to 14229.5] | 8462.9 [6703.2 to 17697] | 7162 [456 to 19814.4] | 16418.5 [5184.5 to 22000] | 3124.1 [615.6 to 7653.1]
  2019-nCoV S/293F-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  2019-nCoV S/293F-1000 at Month 4-Peru | 1159.1 [611.5 to 2272.9] | 12284.6 [7426.9 to 17142.3] | 2039.4 [722.3 to 5816] | 12227.4 [1528 to 19363.6] | 11351.8 [4295.6 to 17359.4] | 20226.2 [12771.2 to 22000] | 11395.5 [4846.1 to 19119.8]
  2019-nCoV S/293F-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 33 | 29 | 45
  2019-nCoV S/293F-1000 at Month 4-Total | 1159.1 [611.5 to 2097.5] | 1027.8 [180.7 to 2376.2] | 1917.6 [638.8 to 5311.8] | 6339.8 [1690.5 to 19297.5] | 8064.2 [2891.2 to 15134.2] | 16315.5 [7446.2 to 21740.8] | 4329.2 [1293.8 to 13465.2]
  2019-nCoV S/293F-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 13 | 13 | 26
  2019-nCoV S/293F-1000 at Month 4-USA | 1182.9 [680.1 to 1756.6] | 206.6 [123.1 to 643.1] | 1867.5 [816.7 to 4612.3] | 2586.8 [1695.2 to 15358.5] | 5671.2 [341 to 8064.2] | 11730.5 [1608.5 to 16981.8] | 1706.6 [993.1 to 4302.8]
  229E-RBD-50 at Month 0-Peru: number analyzed (Participants) | 15 | 4 | 15 | 18 | 19 | 24 | 45
  229E-RBD-50 at Month 0-Peru | 6075 [4465.1 to 7750.2] | 8687.5 [5760.1 to 10086.8] | 4655.5 [4012.8 to 5647.9] | 9766.1 [7655.8 to 13076.6] | 7667.2 [4595.1 to 8742.5] | 8987 [7051.7 to 11952.9] | 5536.8 [4000.8 to 7704.2]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 29 | 19 | 29 | 28 | 35 | 38 | 82
  229E-RBD-50 at Month 0-Total | 4321.2 [2266.5 to 6227] | 3656.5 [1687.5 to 7638.4] | 4164 [3314.8 to 5418.8] | 8399.5 [6223.2 to 10962] | 5609 [2988 to 7861.2] | 7848.9 [5618.9 to 10069.6] | 4889.6 [3536.6 to 7270.6]
  229E-RBD-50 at Month 0-USA: number analyzed (Participants) | 14 | 15 | 14 | 10 | 16 | 14 | 37
  229E-RBD-50 at Month 0-USA | 2664.1 [1670.3 to 4190.9] | 2398.2 [1687.5 to 6818.2] | 3365.1 [2633.3 to 4118.2] | 6920.4 [3539.1 to 7853.8] | 3977.8 [1847.7 to 7549] | 5114.9 [3390.9 to 7718.6] | 4339.2 [2300.5 to 5952]
  229E-RBD-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 18 | 16 | 33
  229E-RBD-50 at Month 2-Peru | 5480.5 [4087 to 7269.6] | 10204.8 [8883.9 to 11525.6] | 5184.4 [4430.1 to 6217.2] | 9299.8 [7956.5 to 12819.2] | 6259.1 [3543.9 to 7812.8] | 9592.9 [8265.1 to 12218.4] | 6666.8 [4642.2 to 8523]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 38 | 36 | 31 | 32 | 76
  229E-RBD-50 at Month 2-Total | 4491 [2831.5 to 6643.6] | 5538.9 [3732.4 to 7727.1] | 4630.2 [3039 to 5985.9] | 7680.6 [4568.6 to 9781.8] | 4738.2 [3038.9 to 7294.2] | 7152.1 [4167.4 to 9633.8] | 4715.8 [2662.9 to 7221.8]
  229E-RBD-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 19 | 13 | 16 | 43
  229E-RBD-50 at Month 2-USA | 2676.5 [1714.2 to 3997.5] | 4896 [3052.1 to 7001] | 3227.9 [2265.4 to 5141.9] | 5982 [2890.2 to 7680.6] | 4185.8 [2660.5 to 5522.2] | 4205.8 [1024.2 to 5512.7] | 3671.8 [2322.8 to 5293.4]
  229E-RBD-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 16 | 14 | 17 | 14 | 16
  229E-RBD-50 at Month 4-Peru | 5674.4 [3985.6 to 6540.4] | 12835.4 [11581.9 to 14088.8] | 6628.8 [5038.1 to 7600.2] | 10900.1 [8523.8 to 13950.5] | 7793 [6289 to 8675] | 11288.1 [9721 to 12000.3] | 6895.5 [5185.4 to 10066.9]
  229E-RBD-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 26 | 24 | 29 | 24 | 40
  229E-RBD-50 at Month 4-Total | 4769.4 [3819.2 to 6273] | 7684.5 [4887.2 to 9870.4] | 5758 [3363.9 to 7464.1] | 8742.8 [6231.1 to 13223.6] | 6800.8 [4781.8 to 8223.5] | 9087.4 [6173.9 to 11392.2] | 5392 [3585.4 to 7818.9]
  229E-RBD-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 10 | 12 | 10 | 24
  229E-RBD-50 at Month 4-USA | 3782.9 [2974.6 to 4094.6] | 5549.1 [4096.2 to 7278.8] | 3770.2 [1311.6 to 5784.1] | 6330 [4810.5 to 9281.8] | 6125 [3926.9 to 7413.3] | 6074.2 [3362.9 to 7725.6] | 4619.6 [2416.6 to 6273.1]
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 25 | 16 | 21 | 44
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru | 19899 [15659 to 22000] | 14867.4 [7324.9 to 22000] | 22000 [18506.6 to 22000] | 14711 [9667.2 to 20261.8] | 21350.2 [13585.1 to 22000] | 14855.8 [10743 to 20445.8] | 10342.2 [7780.1 to 16512.4]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 46 | 37 | 42 | 93
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 17290.1 [9474.8 to 22000] | 8322.4 [5403.6 to 13950.9] | 21138.5 [13965 to 22000] | 15478.8 [9890.9 to 21045.4] | 15729 [8237.5 to 22000] | 14555.8 [7663.9 to 21172.6] | 10404 [6037 to 14504.8]
  HCoV-229E S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 21 | 21 | 21 | 49
  HCoV-229E S1S2 ECD His-50 at Month 0-USA | 10297.5 [5067.8 to 21442.2] | 7937 [4195.2 to 11355.8] | 19071.6 [9260.4 to 22000] | 16298 [10831 to 22000] | 11982.2 [4528.8 to 20300.2] | 11300 [4945.2 to 22000] | 10404 [3929.2 to 13611.8]
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 18 | 16 | 35
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru | 15490 [10239.5 to 21122.4] | 21984.2 [21976.4 to 21992.1] | 13781.4 [11054.8 to 16781.7] | 15861.8 [9562 to 18270.5] | 12104.6 [6711.9 to 16836.2] | 13485.8 [8237.2 to 16891.2] | 7754 [5060.9 to 13578.6]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 35 | 12 | 39 | 36 | 31 | 32 | 78
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 13251.8 [7342.4 to 18761.9] | 7710.4 [5495.2 to 19288.2] | 12450.5 [8284.1 to 16509.5] | 10741.6 [8022.8 to 16222.2] | 10419.2 [7264.8 to 15295.5] | 10632 [5095.2 to 16246.6] | 6951 [4356.9 to 11729]
  HCoV-229E S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 12 | 10 | 19 | 19 | 13 | 16 | 43
  HCoV-229E S1S2 ECD His-50 at Month 2-USA | 7194.9 [1959.9 to 9653] | 7437.2 [5424.6 to 8784.2] | 8613.5 [3376.6 to 14622.9] | 9110.2 [6944.4 to 11406.2] | 9798 [8471.5 to 13046.2] | 6805.5 [1312.6 to 13434.1] | 6789.5 [3251.5 to 9647.5]
  HCoV-229E S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 19 | 14 | 18
  HCoV-229E S1S2 ECD His-50 at Month 4-Peru | 12664 [8975.7 to 17440.9] | 21957.2 [21935.9 to 21978.6] | 12504.6 [7820.4 to 18872.4] | 13619.5 [10011.1 to 16479.2] | 11718 [7236 to 16642.8] | 11386.5 [6412.5 to 14079.9] | 7465.9 [5161.4 to 11797.5]
  HCoV-229E S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 31 | 26 | 43
  HCoV-229E S1S2 ECD His-50 at Month 4-Total | 10593.6 [6351.4 to 15398.7] | 19506.5 [10245 to 21978.6] | 9961.5 [6591.2 to 19333.9] | 12133.1 [8811.9 to 14841.1] | 11396 [6578 to 14176.4] | 11556.8 [6052.5 to 15732.1] | 7501.2 [4611 to 12510.5]
  HCoV-229E S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 12 | 25
  HCoV-229E S1S2 ECD His-50 at Month 4-USA | 6045.6 [4207.4 to 7005.4] | 12529.5 [7219.9 to 18323.9] | 7846.5 [4158.8 to 19113.9] | 9651.5 [6913.8 to 12437.8] | 10991.1 [5297.5 to 13288.2] | 11764.9 [6239.4 to 16624.1] | 7501.2 [2969.8 to 12632.5]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 25 | 16 | 21 | 44
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru | 11668.8 [5203 to 16714] | 15622.9 [10535.9 to 20041.5] | 20251.9 [11690.9 to 22000] | 22000 [12186.2 to 22000] | 17805.8 [10662.1 to 20763.2] | 19896.8 [16454 to 22000] | 15293.1 [9350.9 to 22000]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 46 | 37 | 41 | 93
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 10373.5 [4227.2 to 17610.3] | 11830.1 [7079.6 to 20054.6] | 20251.9 [9224.1 to 22000] | 17539.9 [12178.6 to 22000] | 14465 [9054 to 20689.2] | 19475.8 [14455.2 to 22000] | 14566.8 [7623 to 21648.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 21 | 21 | 20 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA | 7752.8 [2475 to 20000.5] | 10792.8 [4975.6 to 19968.2] | 20279.6 [8633.2 to 22000] | 14482.8 [10836.2 to 19693.2] | 13855.8 [7185 to 19375.8] | 17473.6 [11148.2 to 22000] | 13830.5 [5683.2 to 20382.5]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 18 | 16 | 36
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru | 10629 [7875.9 to 15722.1] | 20287.9 [19431.8 to 21143.9] | 11187 [7741.8 to 22000] | 18858.8 [7010.2 to 22000] | 14461.6 [11335.4 to 20452.8] | 22000 [21078.8 to 22000] | 14260.8 [9801.1 to 19572.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 38 | 36 | 30 | 32 | 79
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 12036.5 [6845 to 17650.2] | 15556 [11395.4 to 21613.9] | 12295.6 [7485.9 to 20675.4] | 14119.9 [7793.1 to 22000] | 13228.8 [6242.9 to 18775.9] | 21639 [11705.7 to 22000] | 13306.2 [8014.2 to 18093.1]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 19 | 12 | 16 | 43
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA | 15608.5 [1507.5 to 19182.2] | 14067.4 [10970.8 to 20364.4] | 13642.8 [7470.8 to 17337.5] | 12119.5 [8763.2 to 18655.6] | 8948.6 [5130.1 to 16518.2] | 12770.5 [7102.8 to 21470.5] | 11295.2 [6278.9 to 16840.4]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 15 | 19
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Peru | 8894.2 [5556.9 to 14511.1] | 22000 [22000 to 22000] | 10096.9 [6855.2 to 15999.6] | 20468.8 [8338.9 to 22000] | 15596.3 [11027.1 to 19896.1] | 17215.8 [12525.4 to 22000] | 15132.5 [9262.5 to 20876.4]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 32 | 28 | 45
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total | 8894.2 [5115.9 to 16139.3] | 16623.1 [9625.1 to 22000] | 10398.2 [6761.2 to 16473] | 16420.5 [8521.2 to 22000] | 15129 [9183.8 to 20451.1] | 16627.8 [10980.5 to 22000] | 12564.5 [7646.8 to 20485.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-USA | 11432.1 [2214 to 21503.7] | 10165.5 [7582.8 to 13934.7] | 10398.2 [6660.2 to 18211.2] | 11051 [8521.2 to 16683.5] | 11546.4 [6935.4 to 20765.9] | 12100.8 [9035.5 to 22000] | 12463.2 [6857.5 to 18039.7]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 24 | 16 | 21 | 45
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru | 1310.2 [1019.5 to 2396] | 807.6 [575.8 to 1401.6] | 1773.8 [408.9 to 3607.5] | 771.4 [1 to 1837.4] | 1 [1 to 1759.4] | 1 [1 to 692.8] | 920.5 [1 to 2928]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 45 | 37 | 42 | 94
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 1652.5 [1033.6 to 2765.2] | 904 [557.1 to 2311.6] | 2163.6 [870.5 to 4423.7] | 1109 [1 to 2274] | 1688.5 [1 to 4138.2] | 1 [1 to 1196.4] | 1302.1 [63.3 to 2763.9]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 21 | 21 | 21 | 49
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA | 2171 [1100.5 to 2829.8] | 904 [369.2 to 2565.6] | 2484.6 [1145.6 to 4467.4] | 2048 [94 to 3609.2] | 3091.2 [422.2 to 4483.8] | 1 [1 to 2562] | 1460.2 [388.5 to 2677.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 21 | 1 | 20 | 16 | 18 | 16 | 31
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru | 2241 [1207.8 to 3753.8] | 5477.8 [5477.8 to 5477.8] | 3263.6 [1880.6 to 4896.8] | 1329.9 [392.9 to 2680.5] | 576.6 [6.5 to 2645.4] | 936.6 [1 to 2939.8] | 658.8 [25.4 to 1771.8]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 29 | 9 | 38 | 35 | 30 | 29 | 69
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 2431.2 [1527.8 to 4081.8] | 1134 [756.5 to 5441.8] | 3725.4 [1644 to 4862.9] | 1474.8 [358.2 to 3332.6] | 1825.9 [480.2 to 4706] | 710.2 [1 to 2920] | 1041.5 [300 to 3206]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 8 | 8 | 18 | 19 | 12 | 13 | 38
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA | 3289.9 [2367.9 to 4426.8] | 1111.6 [742 to 3619.8] | 4343.9 [802.8 to 4765.3] | 2125.8 [393.5 to 3722.8] | 4030.1 [1939.8 to 6035.1] | 201 [1 to 1266.2] | 1885.9 [819.2 to 3440.9]
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 18 | 14 | 18
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Peru | 1418.4 [727.7 to 2977.8] | 2714.9 [2714.2 to 2715.6] | 2002.9 [944.4 to 3543.1] | 1314 [470.6 to 2511.3] | 1372 [677.8 to 1930.9] | 1213.1 [588.2 to 1522.1] | 971.9 [493.4 to 1970.8]
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 30 | 26 | 44
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total | 1370.5 [830.8 to 2874.6] | 1894.6 [721.9 to 2715.6] | 2083.8 [1126.1 to 3673.4] | 1526 [275.3 to 2755.7] | 1561.9 [802.5 to 3617.2] | 1099.9 [343.7 to 2692.8] | 1570 [727.1 to 2633.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 12 | 26
  HCoV-NL63 S1S2 ECD His-50 at Month 4-USA | 1347.5 [1134.4 to 2302.3] | 839.9 [598.9 to 2860.3] | 2242.4 [1261.2 to 4987.2] | 2158 [78.8 to 3082.2] | 3185.5 [968.4 to 4620.1] | 482.2 [209.1 to 3879.1] | 2024.9 [910.7 to 3238.5]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 25 | 16 | 21 | 44
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru | 21654.8 [16901.2 to 22000] | 20565.5 [17515.8 to 22000] | 22000 [22000 to 22000] | 22000 [19747.2 to 22000] | 21985.4 [18529.6 to 22000] | 22000 [20590.8 to 22000] | 22000 [20284.2 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 46 | 37 | 42 | 93
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 21228.5 [11765.6 to 22000] | 22000 [13884.7 to 22000] | 22000 [18979.1 to 22000] | 22000 [16712.6 to 22000] | 21717.8 [16117.5 to 22000] | 22000 [19735.2 to 22000] | 22000 [17619.2 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 21 | 21 | 21 | 49
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA | 20290.5 [10726.8 to 22000] | 22000 [12504.3 to 22000] | 22000 [16110.6 to 22000] | 21400.2 [14904 to 22000] | 20708.5 [14630.8 to 22000] | 21808.2 [19607.5 to 22000] | 22000 [13638.5 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 18 | 16 | 36
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru | 22000 [13788.2 to 22000] | 22000 [22000 to 22000] | 22000 [18316.2 to 22000] | 22000 [12123 to 22000] | 22000 [19496.9 to 22000] | 22000 [22000 to 22000] | 21939.4 [17744.4 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 39 | 36 | 31 | 31 | 79
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 22000 [12979.2 to 22000] | 22000 [21736.1 to 22000] | 22000 [17619.8 to 22000] | 22000 [12700.5 to 22000] | 21747.2 [14016.6 to 22000] | 22000 [21492.6 to 22000] | 22000 [15977.6 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 19 | 19 | 13 | 15 | 43
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA | 22000 [9940.5 to 22000] | 22000 [21208.4 to 22000] | 22000 [15400.6 to 22000] | 22000 [13638.8 to 22000] | 14161.2 [10428.8 to 22000] | 21857.8 [16266.1 to 22000] | 22000 [11849.1 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 15 | 18
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Peru | 17605 [12000.8 to 22000] | 22000 [22000 to 22000] | 16831.6 [13158.9 to 22000] | 22000 [19771 to 22000] | 22000 [19076.5 to 22000] | 22000 [18506.9 to 22000] | 22000 [16550.3 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 32 | 28 | 43
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total | 18049.1 [11269.3 to 22000] | 20167.9 [10548.5 to 22000] | 16831.6 [12711.1 to 22000] | 22000 [17212 to 22000] | 22000 [15154.6 to 22000] | 22000 [17609.3 to 22000] | 22000 [14835.4 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 25
  HCoV-OC43 S1S2 ECD His-50 at Month 4-USA | 19733.5 [7811.6 to 22000] | 13144.2 [7889.9 to 19251.8] | 18198.8 [12508.4 to 22000] | 18645.8 [16707.2 to 22000] | 21096.9 [12738.1 to 22000] | 22000 [16967.2 to 22000] | 22000 [14041.5 to 22000]
  HKU1-RBD-50 at Month 0-Peru: number analyzed (Participants) | 15 | 4 | 16 | 18 | 19 | 24 | 44
  HKU1-RBD-50 at Month 0-Peru | 4680.8 [3475.1 to 8266.1] | 5882.9 [4273.1 to 8219.4] | 4182 [3300.6 to 7167.7] | 6026.9 [3761.6 to 8429.2] | 5722.8 [4614.5 to 8720.2] | 6905.6 [4252.9 to 11249.9] | 4614.2 [2901.8 to 6242.9]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 30 | 19 | 32 | 28 | 34 | 37 | 82
  HKU1-RBD-50 at Month 0-Total | 3685.9 [2425.3 to 4976.2] | 2462.2 [565.8 to 6050.5] | 4182 [3004.1 to 6246.4] | 5345.4 [2956.1 to 8354.8] | 5078.6 [3295.9 to 7475.1] | 5831.5 [3314.8 to 10451.2] | 4299 [2765.1 to 5769]
  HKU1-RBD-50 at Month 0-USA: number analyzed (Participants) | 15 | 15 | 16 | 10 | 15 | 13 | 38
  HKU1-RBD-50 at Month 0-USA | 2414.5 [478.9 to 3875.4] | 967.2 [153.1 to 4143.8] | 4038.2 [2178.6 to 5600.7] | 3248.5 [2614.1 to 5078.7] | 3224 [1979.4 to 5239.5] | 3987.2 [1161.2 to 6409.8] | 4159.8 [2244.8 to 5272.8]
  HKU1-RBD-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 18 | 16 | 33
  HKU1-RBD-50 at Month 2-Peru | 4748.2 [3258.1 to 5663.1] | 9305.6 [7792.4 to 10818.8] | 4049.8 [3332.4 to 5552.1] | 4465.2 [1954.8 to 8036] | 5606.2 [3029.4 to 6972.6] | 8100.4 [6050.7 to 10273.3] | 4642.8 [3140.2 to 5811.5]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 35 | 11 | 38 | 36 | 30 | 32 | 74
  HKU1-RBD-50 at Month 2-Total | 4032 [2750.6 to 5512.5] | 2888 [850.9 to 4814.2] | 3940.1 [2416.6 to 5373] | 4221.2 [1945.1 to 5929.4] | 4755.5 [2264.6 to 6572.6] | 5169 [1606.1 to 8091.3] | 3674.4 [1796.7 to 5306.6]
  HKU1-RBD-50 at Month 2-USA: number analyzed (Participants) | 12 | 9 | 18 | 19 | 12 | 16 | 41
  HKU1-RBD-50 at Month 2-USA | 3937.5 [782.2 to 5200.2] | 2740.8 [803 to 3264] | 3319.1 [1448.1 to 4993.1] | 2854.8 [2050.1 to 4753.5] | 4335.5 [1954.9 to 5833.6] | 1491 [245.3 to 4634.9] | 3182 [1526.2 to 4311.8]
  HKU1-RBD-50 at Month 4-Peru: number analyzed (Participants) | 23 | 2 | 15 | 13 | 17 | 14 | 16
  HKU1-RBD-50 at Month 4-Peru | 4390.2 [2928.5 to 7017.4] | 13067 [12782 to 13352] | 4000.2 [2880 to 5417.9] | 5357.8 [3623.2 to 10625] | 6637.8 [5313.2 to 12187.3] | 8563.5 [5879.8 to 9414.8] | 5364.6 [3907.1 to 7440.5]
  HKU1-RBD-50 at Month 4-Total: number analyzed (Participants) | 31 | 6 | 24 | 24 | 28 | 25 | 38
  HKU1-RBD-50 at Month 4-Total | 3976.5 [2569.6 to 6837.5] | 6590.8 [1939.2 to 11684.8] | 3957.6 [2779.2 to 6059.6] | 5989.2 [3841.5 to 10464.3] | 5765.2 [4747.2 to 9501.9] | 6267 [2413.2 to 8968.5] | 5670 [3024.5 to 7187.1]
  HKU1-RBD-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 9 | 11 | 11 | 11 | 22
  HKU1-RBD-50 at Month 4-USA | 3915.6 [1399.6 to 4973.2] | 2603.9 [1152.1 to 5262] | 3812.2 [601.2 to 7509] | 6620.8 [4232.9 to 9818] | 5373 [3729.4 to 6094.6] | 1736.2 [1209.5 to 5977.9] | 5670 [2819.4 to 6903.2]
  NL63-RBD-50 at Month 0-Peru: number analyzed (Participants) | 15 | 4 | 16 | 18 | 19 | 24 | 46
  NL63-RBD-50 at Month 0-Peru | 14484 [10679.5 to 16088] | 13696.4 [11150.8 to 15540.7] | 13275.8 [10689.8 to 15579.8] | 10680.9 [8479.9 to 17921.4] | 10645 [8987.1 to 15443.4] | 11912.2 [8342.7 to 15520.4] | 14069.2 [10707.1 to 18166.8]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 30 | 19 | 32 | 27 | 35 | 36 | 84
  NL63-RBD-50 at Month 0-Total | 12764.2 [10233.2 to 15747.9] | 9490.5 [4515.8 to 15669.8] | 12702.1 [10038.6 to 15158.8] | 11096.2 [8436.5 to 16162.1] | 11885.5 [8987.1 to 16305.9] | 11120.4 [7035.6 to 14424.9] | 12568.1 [8691.9 to 16769.1]
  NL63-RBD-50 at Month 0-USA: number analyzed (Participants) | 15 | 15 | 16 | 9 | 16 | 12 | 38
  NL63-RBD-50 at Month 0-USA | 11552 [9906.2 to 14993.9] | 9414.2 [3832.9 to 14601.2] | 12460.1 [9466.9 to 14499.1] | 14351.2 [8396.5 to 15247.2] | 12491 [9092.6 to 16777.2] | 8861.4 [4558.1 to 10832.3] | 10617.9 [7594.4 to 15042.6]
  NL63-RBD-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 19 | 16 | 35
  NL63-RBD-50 at Month 2-Peru | 16886.5 [14494.1 to 19482.5] | 19538.5 [18307.8 to 20769.2] | 16900.9 [14757.2 to 19905.1] | 13423.2 [10413 to 16535.8] | 12332 [9137.8 to 17829.5] | 14408.6 [12356.5 to 18697.2] | 15272.5 [10753.6 to 21236.5]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 39 | 36 | 32 | 32 | 78
  NL63-RBD-50 at Month 2-Total | 16187.4 [13743.2 to 19997.6] | 15246.6 [9385.9 to 18307.8] | 15328.8 [11726.8 to 18709.9] | 12649.2 [10162.9 to 16007.6] | 13769.6 [9310.7 to 19473.3] | 11789.5 [7024.7 to 14872.4] | 14403 [9855.5 to 17739]
  NL63-RBD-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 19 | 19 | 13 | 16 | 43
  NL63-RBD-50 at Month 2-USA | 15439 [13683.2 to 20301] | 14859.6 [6395.6 to 15680.6] | 11465.2 [9249.9 to 17730] | 11990 [9580.9 to 14540.6] | 14499.8 [9550 to 20001.8] | 7331.5 [4560 to 10097] | 13760 [8139.9 to 16647.6]
  NL63-RBD-50 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 14 | 19
  NL63-RBD-50 at Month 4-Peru | 16414.2 [14343.3 to 18427.4] | 21475.6 [21213.4 to 21737.8] | 18752.8 [14166.7 to 22000] | 17525 [15082.4 to 19848.1] | 16948.2 [13870.8 to 19255.8] | 15513.4 [13387 to 18576.1] | 17003.2 [15494.2 to 20300.8]
  NL63-RBD-50 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 33 | 27 | 45
  NL63-RBD-50 at Month 4-Total | 16414.2 [14353.2 to 18465.1] | 16318 [6564.5 to 21737.8] | 16138.9 [13322.8 to 21966.8] | 16900.8 [12282.1 to 19721.6] | 17029.5 [13733.5 to 20776.2] | 14393.2 [11098.4 to 17688.4] | 16313.8 [12920 to 18796.2]
  NL63-RBD-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 13 | 13 | 26
  NL63-RBD-50 at Month 4-USA | 16102.8 [15157.6 to 18760.1] | 8271.2 [4730.7 to 14263.6] | 13724.9 [9913 to 16349.1] | 13457.8 [10843.2 to 18114] | 17576.5 [12328.5 to 22000] | 12415 [10593.8 to 16818.2] | 15684.8 [11863.9 to 18141.6]
  OC43-RBD-50 at Month 0-Peru: number analyzed (Participants) | 15 | 4 | 16 | 18 | 19 | 24 | 44
  OC43-RBD-50 at Month 0-Peru | 2985.5 [2566.6 to 4455.9] | 6679.5 [5151.3 to 7903.9] | 3186.8 [2262.6 to 6841.2] | 6486.6 [4237.3 to 10093.1] | 6529.2 [4211.5 to 9933.4] | 6453.1 [3942.5 to 9665.8] | 4586.4 [2770.2 to 6010]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 30 | 19 | 32 | 27 | 34 | 36 | 82
  OC43-RBD-50 at Month 0-Total | 2935.4 [1285.6 to 4766.7] | 5071.2 [2724.9 to 8088.6] | 3162 [2009.2 to 5766.2] | 5100.2 [3351 to 8183] | 4323.4 [3443.5 to 8185.5] | 5370.1 [2853.8 to 9246.1] | 4057.5 [2167.2 to 5839.6]
  OC43-RBD-50 at Month 0-USA: number analyzed (Participants) | 15 | 15 | 16 | 9 | 15 | 12 | 38
  OC43-RBD-50 at Month 0-USA | 1280 [667.8 to 4596.9] | 4605.5 [2724.9 to 7486.6] | 2889 [1456.4 to 5263.1] | 3168.5 [2747.2 to 3803] | 3926 [1839.1 to 4282.2] | 3015.4 [1672.7 to 8357.2] | 3453.2 [1751.2 to 5351.2]
  OC43-RBD-50 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 17 | 17 | 16 | 33
  OC43-RBD-50 at Month 2-Peru | 3673.2 [2494 to 6038] | 8870.6 [8101.7 to 9639.6] | 3561 [1608.7 to 5501.9] | 6385 [5289.5 to 10512.5] | 5122.2 [3203 to 6494.8] | 7340 [4637.5 to 12214.4] | 4977.5 [3439 to 8033]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 38 | 36 | 29 | 32 | 76
  OC43-RBD-50 at Month 2-Total | 3474.9 [2152.3 to 7595.8] | 7070.4 [4944.4 to 10340.4] | 3520.8 [1433.1 to 5827.1] | 5347.4 [3705.7 to 8489.4] | 4034.8 [3186.2 to 6998] | 5495.1 [2247.9 to 10117.6] | 4046 [2388.2 to 5986.6]
  OC43-RBD-50 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 19 | 12 | 16 | 43
  OC43-RBD-50 at Month 2-USA | 2449 [867.5 to 8063.8] | 6665.1 [4109.6 to 9791.8] | 3332 [922.3 to 6568.1] | 3874.2 [2698.1 to 6097.8] | 3852.1 [1810.6 to 7122.4] | 2695.2 [1087.6 to 5851.7] | 3108.5 [1729.2 to 4968.9]
  OC43-RBD-50 at Month 4-Peru: number analyzed (Participants) | 23 | 2 | 15 | 14 | 16 | 14 | 16
  OC43-RBD-50 at Month 4-Peru | 3639.8 [2226.6 to 4428.2] | 12305.6 [11062.2 to 13549.1] | 2662 [1855.8 to 6446.2] | 7468 [5363.2 to 11977.7] | 7015 [4843.3 to 11032.9] | 8543.6 [6634.9 to 11048.1] | 5337 [4809.8 to 8129.5]
  OC43-RBD-50 at Month 4-Total: number analyzed (Participants) | 31 | 6 | 25 | 25 | 27 | 27 | 40
  OC43-RBD-50 at Month 4-Total | 3609.2 [2161.1 to 4428.2] | 4994.5 [3637.4 to 8680.9] | 2662 [1454.8 to 5753.5] | 7003 [4924.5 to 11003.5] | 6118 [4052.6 to 9976.9] | 7069.8 [4899.1 to 11790.6] | 5000.4 [2824.2 to 7358.4]
  OC43-RBD-50 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 11 | 11 | 13 | 24
  OC43-RBD-50 at Month 4-USA | 2245 [2013.6 to 4268] | 3998.8 [2895.9 to 4858] | 2509 [1075.7 to 5299.2] | 6620 [4530 to 7212.1] | 5568.2 [2614.8 to 7064] | 6559.8 [1678.5 to 12224.8] | 3969.9 [2216.8 to 6878.8]
  SARS-CoV-2 DB His-1000 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 DB His-1000 at Month 0-Peru | 2272.1 [1064.8 to 5210.2] | 3001.1 [242.5 to 8888.3] | 8110.5 [1215 to 13445.2] | 12070.2 [5880.1 to 21662.9] | 21820.8 [13643.9 to 22000] | 22000 [21660.5 to 22000] | 12744.2 [4012 to 21697.5]
  SARS-CoV-2 DB His-1000 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 49 | 48 | 50 | 97
  SARS-CoV-2 DB His-1000 at Month 0-Total | 1172.4 [92.1 to 3058.3] | 694.5 [1 to 2723.8] | 4689.5 [1215 to 10569] | 6640.5 [2355.5 to 16510] | 13772.8 [5428.8 to 22000] | 21909.8 [10946.5 to 22000] | 4607.2 [1268.8 to 14735]
  SARS-CoV-2 DB His-1000 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 25 | 48
  SARS-CoV-2 DB His-1000 at Month 0-USA | 162.8 [1 to 1354.6] | 694.5 [1 to 2000.9] | 3478.1 [1517.6 to 6497.4] | 3557.4 [1738.7 to 12147] | 7541.4 [1296.2 to 13560.9] | 14427.5 [4669.8 to 22000] | 1301.9 [412.8 to 4977.8]
  SARS-CoV-2 DB His-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 17 | 22 | 18 | 36
  SARS-CoV-2 DB His-1000 at Month 2-Peru | 705 [467.2 to 1687.2] | 7273.9 [4467.3 to 10080.4] | 1634.2 [291.6 to 2563.8] | 5485.5 [3341.5 to 9169.8] | 8686.4 [1878.1 to 12229.2] | 14203.2 [7380.3 to 22000] | 4075.5 [2237.3 to 10192.5]
  SARS-CoV-2 DB His-1000 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 37 | 39 | 36 | 37 | 78
  SARS-CoV-2 DB His-1000 at Month 2-Total | 634.5 [217.9 to 1528.3] | 676.6 [69.6 to 1921.9] | 1088.8 [373.8 to 2889] | 3341.5 [1056.4 to 7316.1] | 4251.4 [496.8 to 11344] | 6804.8 [2819.2 to 15256.5] | 1694 [553.7 to 4726.6]
  SARS-CoV-2 DB His-1000 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 22 | 14 | 19 | 42
  SARS-CoV-2 DB His-1000 at Month 2-USA | 292.5 [112 to 1246] | 470.9 [23.9 to 939.1] | 842.6 [489.4 to 3606.4] | 1600.8 [941.5 to 5260.6] | 1554.5 [390.1 to 5356.8] | 3858.5 [1356.9 to 7079.5] | 657.8 [182.6 to 2197.5]
  SARS-CoV-2 DB His-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 16 | 19
  SARS-CoV-2 DB His-1000 at Month 4-Peru | 401.9 [291.2 to 694.9] | 4613.4 [2861.3 to 6365.4] | 544.1 [162.6 to 1050.5] | 3231 [218.9 to 5238.8] | 3738.6 [550.9 to 5867.6] | 5318.6 [3252.5 to 11144.8] | 2636.5 [1316.9 to 5056.1]
  SARS-CoV-2 DB His-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 32 | 29 | 45
  SARS-CoV-2 DB His-1000 at Month 4-Total | 380 [226.9 to 653.1] | 223.9 [182.4 to 896.2] | 425.9 [209.8 to 857.4] | 918.1 [279.7 to 5238.5] | 2361.4 [419.9 to 4192.9] | 4971.8 [1490.8 to 7960.8] | 1322.5 [444 to 3621]
  SARS-CoV-2 DB His-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 DB His-1000 at Month 4-USA | 236.1 [154.6 to 386.2] | 185.1 [135.1 to 207.2] | 415.8 [322.5 to 597] | 764.8 [280.8 to 4100.2] | 880.8 [188.6 to 1731.3] | 1522.8 [853.5 to 7447.2] | 536.9 [201.3 to 1507.8]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Peru | 2329.5 [1005.4 to 5028.4] | 1503.4 [298.7 to 5402.8] | 8985.8 [2113.8 to 21986.2] | 15238.5 [6794.8 to 22000] | 22000 [15314.7 to 22000] | 22000 [22000 to 22000] | 8798.8 [2016.5 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 49 | 47 | 50 | 97
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total | 1884 [171 to 4922.2] | 455 [37.4 to 3746.6] | 13842 [2503.8 to 21986.2] | 18167.5 [8253.2 to 22000] | 18282 [9827.1 to 22000] | 22000 [20043.4 to 22000] | 6321.5 [1652.2 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 25 | 48
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-USA | 419 [1 to 3479.5] | 454.6 [4.4 to 3746.6] | 15998 [3160.6 to 21518.5] | 18560 [10265.1 to 22000] | 12634.5 [2476.6 to 22000] | 22000 [17478.2 to 22000] | 4664.8 [768.9 to 20479.6]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 18 | 19 | 22 | 18 | 34
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Peru | 614.8 [392.2 to 772.5] | 3533.1 [2698.9 to 4367.3] | 938.9 [287.9 to 2349.7] | 4508 [1109.4 to 6349.9] | 5677.9 [1321.9 to 18651.1] | 9158.1 [4082.4 to 22000] | 3019.4 [805.6 to 6961]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total: number analyzed (Participants) | 35 | 11 | 35 | 41 | 36 | 36 | 75
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total | 587.8 [337.4 to 1037.4] | 743 [90.9 to 1805.5] | 1485.5 [520.5 to 3719.6] | 5276 [1747 to 9449.2] | 5411.9 [581.4 to 14784.2] | 8853.1 [4646.4 to 14318.2] | 1755.5 [569.2 to 4882.2]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-USA: number analyzed (Participants) | 12 | 9 | 17 | 22 | 14 | 18 | 41
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-USA | 371.1 [197.8 to 1902.9] | 282.5 [80.2 to 944.2] | 3212.2 [1006.8 to 10107.2] | 6872.9 [2322.2 to 15478.2] | 4223.1 [385.2 to 10834] | 7731.5 [5068.4 to 13451.9] | 1301.5 [303.2 to 3673.8]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 13 | 18 | 16 | 17
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Peru | 179.9 [128.4 to 363.2] | 1295.8 [1124 to 1467.5] | 316 [234.1 to 481.1] | 1731.8 [398.8 to 2258] | 1442.9 [320.6 to 3319.8] | 2589.5 [834.2 to 4785.1] | 698.2 [493.8 to 2218.8]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 26 | 30 | 28 | 40
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total | 185.8 [128.4 to 363.2] | 647.2 [267.4 to 1467.5] | 341 [216.4 to 600.2] | 1779.8 [452.7 to 4149.4] | 1122.5 [287.9 to 2978.9] | 1776.8 [507.5 to 4489.2] | 556.9 [377.6 to 1292.9]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 12 | 23
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-USA | 242.9 [161.5 to 1067.7] | 292.4 [215.8 to 815.1] | 443.9 [161.5 to 1044.1] | 2524 [659.2 to 4267.8] | 705 [219.2 to 1810.2] | 833.4 [386.3 to 3992.8] | 422.5 [153.9 to 1011.1]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Peru: number analyzed (Participants) | 14 | 4 | 16 | 17 | 19 | 23 | 47
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Peru | 1226.9 [769.1 to 3342.9] | 782 [56.9 to 3556.8] | 4992.5 [3063.4 to 12338.3] | 11573.2 [5604 to 17840.2] | 18083.2 [15367.6 to 21250.9] | 22000 [14180.9 to 22000] | 14558.5 [3418 to 21907.8]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total: number analyzed (Participants) | 28 | 19 | 32 | 29 | 35 | 38 | 83
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total | 792.2 [1 to 1432.1] | 741.2 [1 to 1349.2] | 3937.5 [2489.8 to 8993.9] | 8441.2 [4226.8 to 16106] | 12012 [8091.1 to 20255.2] | 16904.5 [9754.9 to 22000] | 3888 [1467.2 to 15401.6]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-USA: number analyzed (Participants) | 14 | 15 | 16 | 12 | 16 | 15 | 36
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-USA | 13.4 [1 to 978] | 741.2 [1 to 1179] | 2803.5 [458.7 to 5584.9] | 6295.4 [2100.6 to 10299.3] | 5952.6 [1129.8 to 11072.9] | 10463.5 [5537.5 to 15002.4] | 1830 [413.9 to 3857.4]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 21 | 18 | 36
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Peru | 489.5 [322 to 1176.9] | 7622.2 [4443.2 to 10801.2] | 1177.2 [289.9 to 2273.6] | 3506 [1798.4 to 8417.8] | 7619.2 [1618 to 9419.5] | 15530.8 [10028.8 to 22000] | 4801.1 [2781.6 to 8004.9]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 36 | 41 | 35 | 37 | 78
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total | 434.6 [229 to 1084] | 751.6 [81.8 to 1607.1] | 1330.4 [376 to 2229.9] | 3245.2 [962.5 to 7709.2] | 3188.2 [822.6 to 8989.9] | 9842.2 [3396.5 to 16514] | 1820 [569.8 to 4819.9]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 17 | 22 | 14 | 19 | 42
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-USA | 362.2 [85.5 to 1048.8] | 219.5 [51.8 to 1465] | 1483.5 [496 to 2111.2] | 1922.9 [868 to 6178.5] | 1465.6 [235.3 to 4535.2] | 4840.5 [1480 to 9467.4] | 652.1 [278.1 to 1644.6]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 19 | 16 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Peru | 330.1 [197.5 to 523.5] | 4673.1 [2582.1 to 6764.2] | 353 [235.3 to 1184.1] | 2770.9 [320.4 to 4245.5] | 2815.2 [743.5 to 5771] | 7131.1 [3416.5 to 13282.6] | 3884.2 [1348.5 to 5530.6]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 31 | 29 | 45
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total | 301.8 [182.9 to 485] | 230.4 [72.4 to 443.1] | 384.2 [228.8 to 1249.1] | 1359.2 [318.5 to 4397.5] | 2078 [494.9 to 5331.9] | 5453.2 [2084.5 to 8042.8] | 997.2 [322.2 to 3895.5]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-USA | 272.8 [139.7 to 434.1] | 102 [39.5 to 195.8] | 427.8 [240.4 to 1123.4] | 489 [318.5 to 6099.5] | 1042.9 [134.8 to 1957.4] | 3039 [337.2 to 5453.2] | 382.8 [200.1 to 985.1]
  SARS-CoV-2 S1 C His-1000 at Month 0-Peru: number analyzed (Participants) | 22 | 4 | 25 | 22 | 22 | 25 | 49
  SARS-CoV-2 S1 C His-1000 at Month 0-Peru | 1450.6 [774.5 to 3670.2] | 2351 [153.7 to 8355.9] | 5647.5 [563.8 to 12682.5] | 14945.9 [6303.8 to 22000] | 22000 [14979.6 to 22000] | 22000 [21077.8 to 22000] | 16546 [3766.2 to 22000]
  SARS-CoV-2 S1 C His-1000 at Month 0-Total: number analyzed (Participants) | 46 | 22 | 52 | 45 | 46 | 50 | 97
  SARS-CoV-2 S1 C His-1000 at Month 0-Total | 938.8 [53.6 to 2176.2] | 654.9 [34 to 2352.7] | 3900.2 [563.6 to 7742.9] | 8602.8 [2383.2 to 17571.2] | 14027.5 [3387.9 to 22000] | 22000 [8782 to 22000] | 4251 [895 to 18275.8]
  SARS-CoV-2 S1 C His-1000 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 27 | 23 | 24 | 25 | 48
  SARS-CoV-2 S1 C His-1000 at Month 0-USA | 107.2 [1 to 1106.9] | 654.9 [5.4 to 1677.8] | 3034.5 [954.6 to 6494.1] | 2889.5 [1575.6 to 11238.9] | 7256.8 [1109.3 to 14340.8] | 11397 [5061.5 to 22000] | 1044.6 [290.7 to 4973.8]
  SARS-CoV-2 S1 C His-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 20 | 19 | 22 | 18 | 36
  SARS-CoV-2 S1 C His-1000 at Month 2-Peru | 607.5 [239.2 to 1220.4] | 8367.4 [4913.8 to 11820.9] | 1056.9 [150.6 to 2012.8] | 5299.5 [1063.6 to 8401.8] | 10770.6 [1744.4 to 12486.9] | 16795.2 [7519.1 to 22000] | 5463.8 [1750.4 to 12009.3]
  SARS-CoV-2 S1 C His-1000 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 38 | 41 | 36 | 37 | 77
  SARS-CoV-2 S1 C His-1000 at Month 2-Total | 373.1 [162.6 to 1122.8] | 527.5 [42.1 to 1650.9] | 819.9 [192.5 to 1990.2] | 2153.2 [618 to 6854] | 3908 [231.4 to 11546.8] | 8501.5 [3085.5 to 17745.2] | 1748.8 [368.8 to 5473.2]
  SARS-CoV-2 S1 C His-1000 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 18 | 22 | 14 | 19 | 41
  SARS-CoV-2 S1 C His-1000 at Month 2-USA | 214.5 [86.5 to 771.2] | 220 [33.2 to 1277.4] | 521.6 [214.9 to 1875.2] | 1472.5 [529.2 to 4961.9] | 1453.1 [202.8 to 4516.6] | 4590 [826.6 to 8820.5] | 476.8 [172.5 to 1906]
  SARS-CoV-2 S1 C His-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 15 | 20 | 16 | 19
  SARS-CoV-2 S1 C His-1000 at Month 4-Peru | 330.5 [190.8 to 486.6] | 5505.8 [3170.1 to 7841.4] | 585.1 [131.8 to 719.4] | 4116.8 [309.6 to 5886.4] | 3952.8 [513.6 to 5890.4] | 7362.5 [3965.2 to 12498.9] | 2819.8 [1179.6 to 6570]
  SARS-CoV-2 S1 C His-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 28 | 32 | 29 | 45
  SARS-CoV-2 S1 C His-1000 at Month 4-Total | 252.5 [161.7 to 446.2] | 118.9 [69.1 to 656] | 332.1 [185.2 to 736.7] | 685.4 [262.6 to 5740.9] | 1777.1 [404.9 to 4717.2] | 5922.5 [1578 to 8962.2] | 1062.8 [235.8 to 3485.8]
  SARS-CoV-2 S1 C His-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2 S1 C His-1000 at Month 4-USA | 155.1 [110.4 to 261.3] | 85.1 [46.2 to 118.1] | 299.1 [243.1 to 648.5] | 432.8 [268 to 4739.2] | 994.9 [122.4 to 1886.6] | 1989 [571.2 to 6985.5] | 349.8 [140 to 1144.1]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 25 | 23 | 24 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Peru | 1696.2 [830.9 to 3348.9] | 998.9 [476.2 to 4516.8] | 3486.2 [1476.2 to 11336] | 15417.5 [8476.2 to 22000] | 14651.5 [9520.1 to 22000] | 22000 [18660.2 to 22000] | 13939.8 [6797.8 to 18247.8]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total: number analyzed (Participants) | 47 | 22 | 53 | 49 | 47 | 50 | 97
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total | 885 [94.4 to 2685] | 656.2 [29.2 to 4055.2] | 3887.5 [1278.2 to 9165.5] | 6299.2 [3413 to 17363.8] | 11095 [4335.2 to 15640.6] | 20107.8 [10867.4 to 22000] | 5338.2 [1286.2 to 15321.2]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 23 | 25 | 48
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-USA | 223.5 [24.1 to 1728.4] | 578.5 [25.1 to 4055.2] | 4259.2 [1051.3 to 7644.1] | 5231.5 [2196.2 to 7207.3] | 7229.5 [2171.5 to 11993.9] | 12049 [8752.8 to 22000] | 1919.4 [489 to 4345.4]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Peru: number analyzed (Participants) | 21 | 2 | 19 | 19 | 22 | 17 | 35
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Peru | 494 [238.5 to 909.2] | 10406.2 [5576.9 to 15235.6] | 1474.2 [249.5 to 4132.9] | 4938.2 [2573.2 to 7135.8] | 7757.4 [1805.2 to 13836.7] | 19485.8 [9937.8 to 22000] | 5311.5 [2412.4 to 9359.8]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total: number analyzed (Participants) | 32 | 11 | 36 | 41 | 35 | 36 | 74
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total | 448 [176.4 to 1371.9] | 307 [99.8 to 3736.5] | 1524.2 [258.9 to 3482.9] | 3972.8 [1714.2 to 7157.5] | 3793.2 [1557.4 to 11462.9] | 9353.9 [4380.9 to 19869] | 2243.9 [578.3 to 7630.4]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-USA: number analyzed (Participants) | 11 | 9 | 17 | 22 | 13 | 19 | 39
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-USA | 345 [102 to 1663.4] | 227 [20 to 2668] | 2272.2 [384.8 to 3335] | 3806.2 [1321.6 to 7390.8] | 2130.5 [282 to 6566.5] | 6990.8 [2255 to 9507] | 686.5 [262.8 to 2541.6]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 16 | 13 | 18 | 16 | 17
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Peru | 306.5 [179.9 to 642.4] | 7358.9 [4084.9 to 10632.8] | 457.8 [114.6 to 1290.4] | 2838.8 [515 to 5544.8] | 3457.9 [771.6 to 5238.9] | 5575.5 [3571.1 to 14695.4] | 2745.8 [1451.2 to 7510.5]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 25 | 26 | 30 | 28 | 41
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total | 290.8 [179.9 to 642.4] | 527.8 [72.6 to 2350.4] | 475 [129.8 to 1255] | 2359 [740.4 to 5348.9] | 1877 [376.6 to 4065.7] | 6120 [2953.8 to 9433.5] | 1178 [365.8 to 5440]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 9 | 13 | 12 | 12 | 24
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-USA | 240.9 [168.9 to 643.2] | 129.9 [14.7 to 899.2] | 581.8 [146.5 to 788.8] | 1288 [911.2 to 4761] | 887.2 [43.8 to 2504.4] | 6323.6 [450.1 to 8479.2] | 468.8 [165.2 to 1252.9]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 48
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Peru | 8176.2 [4294.2 to 10606.5] | 5839.9 [2648.2 to 11640.8] | 11742 [6655.5 to 22000] | 22000 [18757 to 22000] | 22000 [20991.6 to 22000] | 22000 [22000 to 22000] | 22000 [13059.6 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 51 | 47 | 50 | 97
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total | 4511.2 [217.2 to 9141] | 3607.8 [74.1 to 9263.8] | 10723.5 [6655.5 to 20231.5] | 18757 [8573.1 to 22000] | 22000 [13948.8 to 22000] | 22000 [22000 to 22000] | 14302.8 [4640.5 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 23 | 25 | 49
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-USA | 716.8 [89.8 to 6154.6] | 3377.6 [50.3 to 9152.7] | 10606.9 [6801.1 to 17332.1] | 9666.2 [6437.3 to 20803.1] | 18665 [5514.1 to 22000] | 22000 [17777.8 to 22000] | 5977.8 [2139 to 14994.8]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 18 | 36
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Peru | 2497.5 [1410.8 to 4421.1] | 13223.1 [8834.7 to 17611.6] | 5731.5 [1412.9 to 9827.2] | 12088.8 [8519.5 to 21955.4] | 21598.4 [7961.6 to 22000] | 22000 [19496.1 to 22000] | 14899.1 [8445 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total: number analyzed (Participants) | 36 | 12 | 36 | 41 | 36 | 37 | 79
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total | 2468.5 [1405.9 to 4912.9] | 2873.5 [144.9 to 8252.7] | 6221.2 [2360.1 to 11443.3] | 10721.8 [5993.8 to 21405.5] | 15706.4 [5884.6 to 22000] | 22000 [11296.2 to 22000] | 7608.2 [2573.4 to 16332.9]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-USA: number analyzed (Participants) | 13 | 10 | 17 | 22 | 14 | 19 | 43
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-USA | 2439.5 [328.2 to 5034.8] | 1141.6 [89.8 to 7117.8] | 8299.5 [2834.5 to 12296] | 8169.6 [5845.6 to 17421.4] | 8241.1 [532.2 to 16940.6] | 18872.8 [6146.2 to 22000] | 3458 [1286.9 to 7968.5]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Peru | 1456.8 [733.6 to 2466.3] | 11985.5 [6978.2 to 16992.8] | 1741.6 [759.3 to 5742.8] | 10768.9 [1315.5 to 17353.1] | 11834.2 [3807 to 14293.9] | 18837.4 [11398.3 to 22000] | 9704 [4758.2 to 15637.2]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 33 | 29 | 45
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total | 1456.8 [743.2 to 2466.3] | 1082.2 [120.4 to 3005.2] | 1741.6 [957.9 to 6495.4] | 7205 [1833.8 to 17340] | 8435.5 [3093 to 14028] | 15269 [6482 to 20152.8] | 4275.5 [1547.2 to 11311.2]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 13 | 13 | 26
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-USA | 1367.2 [794.6 to 2324.9] | 144.8 [75.9 to 982.6] | 2163.5 [1144.5 to 7376.4] | 2799.2 [1952 to 16494.5] | 6531.5 [446.8 to 8313] | 11779.2 [1509.8 to 19080] | 2181.5 [1027.4 to 4241.5]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Peru: number analyzed (Participants) | 14 | 4 | 16 | 17 | 19 | 24 | 48
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Peru | 876 [555.5 to 3668.3] | 2067.1 [1079.1 to 7522.2] | 5064.2 [1398.3 to 10949.6] | 22000 [4838 to 22000] | 22000 [17183.5 to 22000] | 22000 [17550.5 to 22000] | 17893.5 [3567.6 to 22000]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total: number analyzed (Participants) | 28 | 19 | 32 | 30 | 35 | 39 | 85
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total | 473.4 [1 to 1547.2] | 140.8 [2 to 914.5] | 2349 [596.8 to 8934.9] | 11627.8 [1568.9 to 22000] | 19478.5 [6490 to 22000] | 20787.5 [5290.9 to 22000] | 4985.5 [1191 to 20774.8]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-USA: number analyzed (Participants) | 14 | 15 | 16 | 13 | 16 | 15 | 37
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-USA | 9.1 [1 to 328.8] | 8.5 [1.2 to 545.8] | 788 [212.9 to 5181] | 3362.2 [869.2 to 12886.8] | 8365.2 [1114.6 to 17173.1] | 5221 [3770 to 16935.6] | 1799.8 [222.5 to 3423.8]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Peru: number analyzed (Participants) | 23 | 2 | 19 | 19 | 22 | 17 | 36
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Peru | 102.2 [56.6 to 429] | 7824.5 [4566.2 to 11082.8] | 685.2 [31.4 to 1508.8] | 3683 [516.2 to 6296.1] | 6996.1 [1120.9 to 15024.8] | 16491.5 [11508.5 to 22000] | 3668.7 [986.3 to 10759.5]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total: number analyzed (Participants) | 35 | 12 | 37 | 41 | 35 | 34 | 75
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total | 92.2 [14.2 to 348.5] | 256.2 [2.8 to 999.9] | 609.8 [46.5 to 1413.8] | 1884.2 [417.5 to 6870.8] | 2501.5 [372.5 to 10071.8] | 7602.9 [1896.7 to 16594.1] | 794.2 [95.6 to 4681]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-USA: number analyzed (Participants) | 12 | 10 | 18 | 22 | 13 | 17 | 39
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-USA | 14.2 [6.6 to 199.2] | 63.9 [1.8 to 422.9] | 413.4 [106 to 1092.7] | 1024.8 [383.2 to 6003.1] | 740.5 [8.2 to 2053.2] | 2081.8 [564.8 to 5172] | 163.5 [17.6 to 746.1]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Peru: number analyzed (Participants) | 24 | 2 | 18 | 16 | 20 | 16 | 19
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Peru | 44.7 [20.8 to 130.9] | 2720.8 [1644.2 to 3797.2] | 224.4 [22.8 to 461.4] | 1209 [53.9 to 2730.4] | 2275.2 [183.4 to 3635.8] | 4180.9 [2490.8 to 7229.2] | 1242 [491.9 to 5010.1]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total: number analyzed (Participants) | 32 | 6 | 28 | 29 | 32 | 29 | 45
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total | 44.4 [20 to 129.5] | 162.6 [1.1 to 506.8] | 183.2 [17.6 to 380.3] | 458.8 [69.8 to 2669.5] | 795.4 [80.1 to 2955.9] | 2540.2 [759.5 to 5222] | 371.5 [46 to 1798.5]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-USA: number analyzed (Participants) | 8 | 4 | 10 | 13 | 12 | 13 | 26
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-USA | 34.9 [14.1 to 93.1] | 1.1 [1 to 81.9] | 101.9 [14.2 to 191.7] | 245.2 [94 to 2669.5] | 344.9 [9.9 to 946.6] | 1035 [99.5 to 2058] | 93.2 [12.1 to 350.4]

3. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (BAMA IgG3) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarizedSARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 24 | 24 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Peru | 22 | 3 | 22 | 21 | 23 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 50 | 48 | 49 | 98
  2019-nCoV S/293F-50 at Month 0-Total | 37 | 13 | 50 | 46 | 44 | 47 | 93
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  2019-nCoV S/293F-50 at Month 0-USA | 15 | 10 | 28 | 25 | 21 | 22 | 44
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Peru | 0 | 0 | 9 | 2 | 12 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  2019-nCoV S/293F-50 at Month 2-Total | 3 | 1 | 23 | 16 | 18 | 6 | 16
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  2019-nCoV S/293F-50 at Month 2-USA | 3 | 1 | 14 | 14 | 6 | 4 | 15
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2 DB His-50 at Month 0-Peru | 22 | 2 | 20 | 17 | 22 | 24 | 47
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2 DB His-50 at Month 0-Total | 32 | 9 | 46 | 40 | 42 | 45 | 81
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 DB His-50 at Month 0-USA | 10 | 7 | 26 | 23 | 20 | 21 | 34
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 DB His-50 at Month 2-Peru | 0 | 0 | 2 | 2 | 8 | 1 | 1
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 DB His-50 at Month 2-Total | 2 | 0 | 12 | 8 | 13 | 2 | 8
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 DB His-50 at Month 2-USA | 2 | 0 | 10 | 6 | 5 | 1 | 7
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 23 | 3 | 23 | 20 | 22 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 41 | 13 | 51 | 44 | 43 | 47 | 96
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 18 | 10 | 28 | 24 | 21 | 22 | 46
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 0 | 0 | 6 | 2 | 11 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 3 | 1 | 20 | 15 | 16 | 6 | 15
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 3 | 1 | 14 | 13 | 5 | 4 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 22 | 24 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 20 | 3 | 22 | 17 | 22 | 25 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 48 | 48 | 49 | 99
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 28 | 10 | 48 | 41 | 41 | 47 | 88
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 8 | 7 | 26 | 24 | 19 | 22 | 39
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 0 | 0 | 4 | 2 | 10 | 1 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 3 | 0 | 14 | 11 | 15 | 5 | 9
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 3 | 0 | 10 | 9 | 5 | 4 | 8
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 22 | 3 | 19 | 19 | 22 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 48 | 49 | 99
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 33 | 11 | 46 | 42 | 42 | 47 | 86
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 11 | 8 | 27 | 23 | 20 | 22 | 37
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 0 | 0 | 4 | 2 | 10 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 3 | 0 | 14 | 13 | 15 | 6 | 9
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 3 | 0 | 10 | 11 | 5 | 4 | 8
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 23 | 3 | 21 | 21 | 22 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 50 | 48 | 49 | 98
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 39 | 14 | 49 | 47 | 43 | 48 | 93
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 23 | 18 | 28 | 26 | 24 | 24 | 48
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 16 | 11 | 28 | 26 | 21 | 23 | 43
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 0 | 0 | 10 | 2 | 14 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 3 | 1 | 26 | 16 | 19 | 6 | 18
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 3 | 1 | 16 | 14 | 5 | 4 | 17
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 22 | 3 | 23 | 21 | 23 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 48 | 49 | 99
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 36 | 13 | 51 | 46 | 44 | 47 | 94
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 14 | 10 | 28 | 25 | 21 | 22 | 44
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 0 | 0 | 7 | 2 | 13 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 3 | 1 | 21 | 16 | 19 | 6 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 3 | 1 | 14 | 14 | 6 | 4 | 13
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 22 | 3 | 20 | 19 | 22 | 25 | 50
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 33 | 11 | 47 | 42 | 42 | 46 | 89
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 11 | 8 | 27 | 23 | 20 | 21 | 39
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 0 | 0 | 8 | 2 | 12 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 3 | 1 | 21 | 15 | 18 | 6 | 12
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 3 | 1 | 13 | 13 | 6 | 4 | 11

4. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (BAMA IgG3) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarizedSARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
MFI
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 24 | 24 | 24 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Peru | 4377 [2471.8 to 8394.2] | 7774.2 [5560 to 10312.6] | 6265.9 [2470.4 to 10721.7] | 5985.4 [2062.8 to 11245.5] | 9181.5 [5618.2 to 12658.5] | 12261.8 [8197.5 to 17973] | 6745.2 [4181.8 to 15152]
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 52 | 50 | 48 | 49 | 98
  2019-nCoV S/293F-50 at Month 0-Total | 2775.6 [406.1 to 6192.9] | 2438.5 [8.6 to 7641] | 6082.5 [3354.8 to 9443.8] | 6652.8 [3177.3 to 12608.7] | 10695.2 [5466.9 to 18239.3] | 11434 [6861.5 to 16712.8] | 5657.4 [3352.8 to 11538.8]
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  2019-nCoV S/293F-50 at Month 0-USA | 1045.5 [207.8 to 2955.5] | 991.6 [8.6 to 5058.5] | 6082.5 [3561.6 to 8754.6] | 7411.9 [4118.8 to 12608.7] | 14983.4 [5466.9 to 21413.5] | 9738.9 [6336.3 to 13702.1] | 5248 [2353.5 to 8077.5]
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Peru |  |  | 622.8 [377.8 to 1412] | 7904.8 [3952.9 to 12097.2] | 2597 [1484.2 to 3392.2] | 2632.5 [2031.9 to 3233.1] | 4400.5 [4400.5 to 4400.5]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  2019-nCoV S/293F-50 at Month 2-Total | 3472.5 [2581.5 to 3573.2] | 11872.5 [11872.5 to 11872.5] | 3146.2 [595 to 4352.5] | 3713 [1790.4 to 7475.8] | 2880 [1484.2 to 4996.9] | 3717.9 [3572 to 4421.4] | 1836.4 [648.1 to 4331.9]
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  2019-nCoV S/293F-50 at Month 2-USA | 3472.5 [2581.5 to 3573.2] | 11872.5 [11872.5 to 11872.5] | 3563.6 [2836.3 to 5393.4] | 3415 [1913.2 to 5502.5] | 5908.8 [2160.2 to 8574.5] | 4109.6 [3592 to 5001] | 1737.2 [581.1 to 4073.9]
  229E-RBD-50 at Month 0-Peru: number analyzed (Participants) | 23 | 3 | 25 | 24 | 24 | 25 | 50
  229E-RBD-50 at Month 0-Peru | 343 [131 to 408.2] | 357.8 [179.4 to 544.4] | 262.5 [115 to 438.2] | 204.9 [2.1 to 430.8] | 233.6 [87.8 to 403.2] | 221 [81.5 to 428] | 322.6 [1 to 606.6]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 47 | 20 | 53 | 49 | 46 | 48 | 95
  229E-RBD-50 at Month 0-Total | 207.5 [12.6 to 384.5] | 49 [1 to 451.1] | 262.5 [84.8 to 456.2] | 224.2 [65.5 to 558] | 256.8 [50.9 to 628.9] | 245 [44.4 to 524.8] | 273.5 [40.2 to 586.5]
  229E-RBD-50 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 28 | 25 | 22 | 23 | 45
  229E-RBD-50 at Month 0-USA | 71.1 [1 to 227] | 1 [1 to 290.8] | 244.2 [72.9 to 463.4] | 268.2 [134.2 to 696.2] | 360.9 [18.3 to 688.8] | 336.2 [41.1 to 531.2] | 230.8 [98.2 to 513]
  229E-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  229E-RBD-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 3.5] | 1 [1 to 1] | 1 [1 to 1] | 181 [181 to 181]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 17 | 23 | 6 | 20
  229E-RBD-50 at Month 2-Total | 16.8 [8.9 to 31.9] | 1 [1 to 1] | 1 [1 to 61.8] | 1 [1 to 6] | 1 [1 to 10.4] | 1 [1 to 1] | 1 [1 to 34.3]
  229E-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 14 | 8 | 4 | 19
  229E-RBD-50 at Month 2-USA | 16.8 [8.9 to 31.9] | 1 [1 to 1] | 1 [1 to 182] | 1 [1 to 292.9] | 1 [1 to 267.9] | 1 [1 to 1] | 1 [1 to 10.4]
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 24 | 50
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru | 21.2 [1 to 61.8] | 335.9 [215.7 to 425.6] | 41.8 [13.8 to 116.8] | 1 [1 to 12.9] | 21.1 [1 to 58.8] | 1 [1 to 1] | 1 [1 to 120.8]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 47 | 48 | 99
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 28.2 [1 to 74.5] | 61 [1 to 330.2] | 47.5 [1 to 148] | 1 [1 to 66.7] | 22.8 [1 to 64] | 1 [1 to 1] | 1 [1 to 98]
  HCoV-229E S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 24 | 49
  HCoV-229E S1S2 ECD His-50 at Month 0-USA | 33.5 [1 to 75.5] | 42 [1 to 159.2] | 68.9 [1 to 158.9] | 16.6 [1 to 446.1] | 22.8 [1 to 119.6] | 1 [1 to 2.1] | 9 [1 to 69]
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 147.2 [74.1 to 388.8] | 4066.5 [4066.5 to 4066.5] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 8.1]
  HCoV-229E S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-229E S1S2 ECD His-50 at Month 2-USA | 147.2 [74.1 to 388.8] | 4066.5 [4066.5 to 4066.5] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 420] | 1 [1 to 15.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 25 | 24 | 24 | 25 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru | 202.8 [102.2 to 358.8] | 742.8 [371.9 to 2045.8] | 397.5 [156 to 499] | 183 [3.8 to 350.2] | 323.9 [221.2 to 611.8] | 232 [113.5 to 485.5] | 403.5 [1 to 1390.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 50 | 47 | 48 | 98
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 268.5 [110.8 to 448.4] | 217 [52.2 to 819.5] | 435.2 [158.2 to 723.2] | 340.5 [146.8 to 1542.7] | 594.5 [274.6 to 1778] | 273 [121.6 to 984.4] | 500.8 [62.5 to 1538.1]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 23 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA | 300.5 [143.8 to 718.8] | 171.2 [52.5 to 726.4] | 463.9 [182.2 to 2537.8] | 918.6 [244.7 to 3551.6] | 1468.8 [602.1 to 2759.2] | 557.2 [150.1 to 1658.5] | 546.5 [147.2 to 1578.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru |  |  | 160.2 [29 to 306.5] | 1 [1 to 1] | 1 [1 to 105.1] | 612.5 [377.4 to 847.6] | 562.2 [562.2 to 562.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 406.8 [276.8 to 626.8] | 8733.2 [8733.2 to 8733.2] | 273.5 [29 to 652.8] | 18.4 [1 to 242.8] | 100.5 [1 to 738.2] | 102.6 [16.5 to 163.2] | 453.1 [127.1 to 1195.1]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA | 406.8 [276.8 to 626.8] | 8733.2 [8733.2 to 8733.2] | 481.5 [22 to 2138.9] | 73.8 [1 to 755.2] | 1350.6 [274 to 3450.6] | 32 [1 to 89.8] | 403.5 [104.1 to 1205.1]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 24 | 50
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru | 4.5 [1 to 38] | 73.6 [1 to 447.8] | 21.2 [1 to 41.5] | 1 [1 to 1] | 1 [1 to 33.4] | 1 [1 to 1] | 1 [1 to 59]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 47 | 48 | 99
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 5.8 [1 to 42.9] | 19.9 [1 to 54.1] | 21.2 [1 to 74.5] | 1 [1 to 48.3] | 1 [1 to 98.2] | 1 [1 to 1] | 1 [1 to 50.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 24 | 49
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA | 7.2 [1 to 63.2] | 19.9 [1 to 50.2] | 20.6 [1 to 83.3] | 1.2 [1 to 302.6] | 32 [1 to 281.5] | 1 [1 to 1] | 1 [1 to 29.8]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 1 [1 to 15.4] | 3743.2 [3743.2 to 3743.2] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA | 1 [1 to 15.4] | 3743.2 [3743.2 to 3743.2] | 1 [1 to 50.1] | 1 [1 to 1] | 1 [1 to 33.8] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 25 | 24 | 24 | 25 | 50
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru | 331 [185.8 to 821.8] | 519.8 [260.4 to 3885.5] | 410.8 [249.5 to 714] | 121.9 [1 to 355.3] | 370.6 [211.7 to 1060.1] | 113.2 [1 to 653] | 364.5 [1 to 1230.7]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 50 | 47 | 48 | 99
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 553.5 [188.1 to 1425.4] | 921.5 [93 to 2026.2] | 581 [249.5 to 1802.2] | 259.8 [72.1 to 2326] | 887 [266.2 to 1540.6] | 359.9 [98.2 to 1018.8] | 485.2 [1 to 2040.5]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 23 | 23 | 49
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA | 618.2 [221.5 to 1736.8] | 932.8 [96 to 1914.9] | 1089.2 [266.4 to 3798.4] | 787 [168.7 to 6205.8] | 1264.2 [604.5 to 7354.4] | 616 [225 to 4806.2] | 967 [131 to 3628.8]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 12 | 3 | 15 | 2 | 1
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru |  |  | 124.5 [3.8 to 269.2] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 519.8 [519.8 to 519.8]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 28 | 18 | 22 | 6 | 20
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 577.5 [552.9 to 802.8] | 22000 [22000 to 22000] | 124.5 [1 to 423.8] | 1 [1 to 1] | 1 [1 to 255.2] | 1 [1 to 1] | 534.5 [7.9 to 1205.4]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 7 | 4 | 19
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA | 577.5 [552.9 to 802.8] | 22000 [22000 to 22000] | 132.5 [1 to 2458.5] | 1 [1 to 41.2] | 272.5 [251.4 to 5251.8] | 1 [1 to 32.6] | 549.2 [5.6 to 1431.8]
  HKU1-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 24 | 24 | 24 | 25 | 47
  HKU1-RBD-50 at Month 0-Peru | 214.2 [75 to 390.2] | 312.8 [156.9 to 366.8] | 212.8 [131.9 to 247.9] | 93.4 [10.6 to 280.9] | 180.8 [104.3 to 372] | 177.8 [1 to 311.5] | 278 [1 to 553.6]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 52 | 50 | 45 | 49 | 95
  HKU1-RBD-50 at Month 0-Total | 146 [42.6 to 305.9] | 39 [1 to 420.8] | 205 [114.1 to 295.8] | 176.2 [40.5 to 328.9] | 188.2 [63.2 to 462.5] | 204 [28.8 to 365] | 230.5 [56.6 to 525.5]
  HKU1-RBD-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 21 | 24 | 48
  HKU1-RBD-50 at Month 0-USA | 121.8 [30 to 267.2] | 20 [1 to 458.2] | 156.6 [99.9 to 420] | 188 [153.7 to 420.4] | 203.8 [33.2 to 513.8] | 255.2 [41.9 to 387.1] | 207.4 [112.9 to 315.4]
  HKU1-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HKU1-RBD-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 49.6] | 1 [1 to 1] | 103 [103 to 103]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HKU1-RBD-50 at Month 2-Total | 131.8 [66.4 to 167.9] | 1 [1 to 1] | 1 [1 to 55.8] | 1 [1 to 1] | 1 [1 to 87] | 1 [1 to 1] | 1 [1 to 108]
  HKU1-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HKU1-RBD-50 at Month 2-USA | 131.8 [66.4 to 167.9] | 1 [1 to 1] | 1 [1 to 106.9] | 1 [1 to 283] | 8.1 [1 to 385.4] | 1 [1 to 48.8] | 1 [1 to 62]
  NL63-RBD-50 at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 22 | 22 | 21 | 25 | 48
  NL63-RBD-50 at Month 0-Peru | 288.8 [38.4 to 480.1] | 497.6 [363.2 to 818.6] | 132.8 [32.6 to 315.4] | 157.1 [1 to 504.4] | 275.5 [80.2 to 505.2] | 243.8 [85 to 413.2] | 194.6 [51.4 to 392.3]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 46 | 20 | 49 | 48 | 43 | 47 | 93
  NL63-RBD-50 at Month 0-Total | 250.1 [3.2 to 386.8] | 14.9 [1 to 406.9] | 178.2 [35.2 to 401.2] | 216.8 [22.4 to 540.8] | 257 [33.9 to 518.4] | 263 [34.8 to 423.1] | 203.8 [24.2 to 408.2]
  NL63-RBD-50 at Month 0-USA: number analyzed (Participants) | 23 | 16 | 27 | 26 | 22 | 22 | 45
  NL63-RBD-50 at Month 0-USA | 154.2 [1 to 377.5] | 1 [1 to 188] | 313 [119.4 to 538] | 279.1 [144.7 to 583.3] | 179.8 [1 to 590] | 304.9 [13.5 to 522.8] | 246.5 [21.8 to 497.2]
  NL63-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  NL63-RBD-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 81.8 [81.8 to 81.8]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  NL63-RBD-50 at Month 2-Total | 122.5 [61.8 to 137.5] | 1 [1 to 1] | 1 [1 to 76.2] | 1 [1 to 161.3] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 12.2]
  NL63-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  NL63-RBD-50 at Month 2-USA | 122.5 [61.8 to 137.5] | 1 [1 to 1] | 1 [1 to 111.1] | 1 [1 to 269.1] | 1 [1 to 125] | 1 [1 to 207.1] | 1 [1 to 6.1]
  OC43-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 25 | 24 | 24 | 24 | 49
  OC43-RBD-50 at Month 0-Peru | 167 [27.5 to 359.5] | 240 [120.5 to 281.8] | 181 [32 to 302] | 132.1 [34.6 to 226.4] | 190.4 [10.8 to 299.6] | 159.8 [60.3 to 437.9] | 156 [1 to 461.2]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 49 | 21 | 53 | 50 | 47 | 48 | 96
  OC43-RBD-50 at Month 0-Total | 110.2 [1 to 254.5] | 101.5 [1 to 323.5] | 157 [1 to 298.8] | 132.1 [24.6 to 311.9] | 149.8 [1 to 478.1] | 189 [35.3 to 379.9] | 154.1 [1.2 to 465.9]
  OC43-RBD-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 23 | 24 | 47
  OC43-RBD-50 at Month 0-USA | 81.4 [1 to 212.6] | 100 [6.2 to 573.8] | 75 [1 to 234.9] | 136.2 [19.9 to 457.1] | 103 [1 to 568.8] | 223.2 [9.4 to 348.5] | 147 [8.6 to 467.9]
  OC43-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  OC43-RBD-50 at Month 2-Peru |  |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 64.5 [64.5 to 64.5]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  OC43-RBD-50 at Month 2-Total | 4.5 [2.8 to 27.5] | 1 [1 to 1] | 1 [1 to 10] | 1 [1 to 107.5] | 1 [1 to 8.9] | 1 [1 to 1] | 1 [1 to 36.1]
  OC43-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  OC43-RBD-50 at Month 2-USA | 4.5 [2.8 to 27.5] | 1 [1 to 1] | 1 [1 to 20.8] | 1 [1 to 162.1] | 1 [1 to 67] | 1 [1 to 12.9] | 1 [1 to 23.9]
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 3 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2 DB His-50 at Month 0-Peru | 1247.8 [659.8 to 2080] | 2987.2 [1494.1 to 4597.2] | 1896.2 [905.2 to 3023.5] | 2111.2 [574 to 4108.2] | 3152.4 [1396.4 to 4115.6] | 3438.8 [1941 to 5054.5] | 2317.4 [1096.1 to 4969]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2 DB His-50 at Month 0-Total | 764.4 [252.4 to 1785.1] | 108.2 [1 to 1962.5] | 1896.2 [912.2 to 3081.2] | 2111.2 [865.8 to 3609.8] | 3284.6 [1267.8 to 5261.2] | 3438.8 [1941 to 5054.5] | 1580 [624.9 to 4279.6]
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 DB His-50 at Month 0-USA | 290 [58.2 to 869] | 96 [1 to 1342.1] | 1883.4 [1010.7 to 3113.5] | 1893.5 [1162.8 to 2980.1] | 4810.2 [1267.8 to 7371.3] | 3307 [2054.8 to 4990.4] | 872.8 [275 to 2740]
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 DB His-50 at Month 2-Peru |  |  | 46.5 [16.5 to 171.2] | 3266.5 [1633.8 to 4457.9] | 494.2 [10.2 to 1133.9] | 465.5 [249.5 to 681.5] | 496.8 [496.8 to 496.8]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 DB His-50 at Month 2-Total | 514.2 [413.9 to 954] | 346.5 [346.5 to 346.5] | 171.2 [3.8 to 717.8] | 312.8 [6 to 1494.4] | 645.2 [10.2 to 1524.4] | 17.2 [1 to 681.5] | 15.4 [1 to 676.1]
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 DB His-50 at Month 2-USA | 514.2 [413.9 to 954] | 346.5 [346.5 to 346.5] | 697.2 [3.1 to 1342.4] | 205.8 [11 to 1201.1] | 1351 [43.4 to 2304.1] | 1 [1 to 341.3] | 9.2 [1 to 696.6]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 4540 [1557 to 8570.2] | 8121.9 [5061.2 to 9750.1] | 6731.5 [1961.8 to 11736.8] | 5331.8 [2050.6 to 6125] | 10606.9 [6633 to 17674.9] | 12610.5 [8540.8 to 20633.8] | 8297.1 [3853 to 14525.3]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 3345.2 [604.8 to 8570.2] | 3968.6 [82 to 9199.1] | 7088.5 [3108.5 to 12626.8] | 7420 [5062.5 to 15174.8] | 12102.8 [6388.2 to 22000] | 13097.5 [7045.8 to 20633.8] | 6348.5 [3134.8 to 11790.8]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 1013.5 [351.1 to 8565.4] | 2257.6 [82 to 8092.4] | 7385.8 [4077.6 to 14141.1] | 10450.8 [8539.1 to 20967.1] | 13650.9 [4723.1 to 22000] | 13518.8 [5902.8 to 19489.2] | 4659 [2641.2 to 9487.2]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru |  |  | 288.5 [207.2 to 1246.8] | 4660 [2330.5 to 13330] | 1506 [403.9 to 2825.5] | 757.8 [742.1 to 773.4] | 2547.2 [2547.2 to 2547.2]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 1482.5 [1187.4 to 5246.1] | 7057.8 [7057.8 to 7057.8] | 1269.5 [274.8 to 3284.2] | 3317.9 [1500.3 to 4612.6] | 1506 [165.9 to 3244.4] | 2865.2 [973.1 to 4958.6] | 1260.2 [336.9 to 2759.6]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 1482.5 [1187.4 to 5246.1] | 7057.8 [7057.8 to 7057.8] | 2885.2 [1281.4 to 5245.7] | 3037.5 [1596.1 to 4345.5] | 1932.1 [1 to 3230.2] | 4707.4 [3535.1 to 5445.4] | 1135 [306.6 to 2956.9]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 22 | 24 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 799.2 [448.3 to 1883.4] | 2001.1 [1428.2 to 3307.8] | 1523.2 [579.2 to 2439.8] | 1568.4 [269.6 to 5099.3] | 2848.6 [1612.4 to 4861.2] | 4569 [2166.5 to 6604.8] | 2606.2 [982.4 to 5748.4]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 48 | 48 | 49 | 99
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 499.6 [114.2 to 1122.8] | 76.5 [4.2 to 1948.2] | 1421.2 [712 to 2314.8] | 2088.5 [579 to 4415.8] | 3197 [1477.4 to 5996.5] | 4066.8 [2331.8 to 6157.2] | 1472.2 [555.9 to 4452.6]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 128.6 [88.1 to 804.4] | 58.5 [4.2 to 1496.1] | 1406 [720.2 to 1990.6] | 2262.2 [880.2 to 3596.2] | 3871.9 [1314.5 to 6343] | 3179.2 [2387.8 to 5427.3] | 780.5 [302 to 2039.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru |  |  | 45.2 [1 to 246.5] | 1562 [781.5 to 2860.5] | 441.8 [51.2 to 1069.8] | 672.8 [432.6 to 912.9] | 1590 [1590 to 1590]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 610.2 [551 to 700.1] | 134 [134 to 134] | 149 [1 to 565] | 980.5 [120 to 2519.4] | 441.8 [1 to 1290.2] | 869 [420.2 to 1019.3] | 173 [1 to 989.9]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 610.2 [551 to 700.1] | 134 [134 to 134] | 431.6 [1 to 826.2] | 959 [131.5 to 1959.9] | 822.4 [1 to 2244.6] | 869 [654.6 to 983.9] | 143.2 [1 to 760.5]
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 1190.8 [693.5 to 1905.8] | 2553.5 [1776.8 to 4001.2] | 1480.2 [578 to 3166.2] | 2077.6 [327.2 to 5539.8] | 3030 [1712.8 to 4956.4] | 4704.8 [2374.2 to 7462.5] | 2987.1 [1258.6 to 6831.9]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 48 | 49 | 99
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 644.6 [170.6 to 1385.9] | 195.2 [3 to 1890.2] | 1595.8 [710 to 2696] | 1709.9 [769.2 to 4666.6] | 3347.6 [1284.1 to 6429.8] | 4140.5 [2164.5 to 6077.8] | 1960.5 [680 to 4877.5]
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 206.2 [98.8 to 580.8] | 107.6 [3 to 770.5] | 1621.8 [754.8 to 2662.4] | 1439.8 [867.5 to 3042.4] | 4387.2 [1139 to 8450.7] | 3513.9 [2124.4 to 5082.6] | 886 [239.2 to 2624.2]
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Peru |  |  | 112.5 [27.5 to 274.2] | 3691 [1846 to 4663.1] | 781.2 [14.5 to 1423.4] | 1147.1 [780.7 to 1513.6] | 1553.8 [1553.8 to 1553.8]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 489.8 [421.1 to 984.6] | 28.8 [28.8 to 28.8] | 205.2 [56 to 957] | 825.1 [136.5 to 1760.3] | 781.2 [14.5 to 1783.6] | 936.4 [669.9 to 1531.7] | 197.2 [1 to 1189.1]
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 489.8 [421.1 to 984.6] | 28.8 [28.8 to 28.8] | 843.5 [146.9 to 1256.4] | 616 [166.8 to 1363.1] | 1355.4 [58.8 to 3433] | 936.4 [703.8 to 1278.6] | 177 [1 to 1161.2]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 6430.5 [3013.2 to 11019.5] | 10084.8 [4316.9 to 16310.5] | 5864 [3558.8 to 12139.2] | 8299 [3134.2 to 22000] | 9396.2 [5386.7 to 17049.7] | 18159 [11974.5 to 21673.8] | 10162.9 [5466.2 to 21283.8]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 48 | 22 | 53 | 50 | 48 | 49 | 98
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 4036.2 [1105.4 to 9311.7] | 6061.8 [109.8 to 10656.9] | 6036.2 [3810 to 10591] | 8299 [3412.7 to 22000] | 14250.9 [6001.6 to 22000] | 16390 [7880.5 to 22000] | 8674.1 [4608.1 to 19279.2]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 23 | 18 | 28 | 26 | 24 | 24 | 48
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 1902.2 [410 to 4706.2] | 4475.5 [109.8 to 10595.1] | 6749.1 [3941.9 to 10170.9] | 8291.6 [4321.6 to 21521.4] | 20010.5 [8572.8 to 22000] | 9598.5 [6330.3 to 22000] | 7004.2 [3149.2 to 15619.1]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru |  |  | 2205 [731.5 to 3424.2] | 5818.5 [2909.8 to 12104.4] | 2566.2 [1860.1 to 5217.4] | 6808.2 [5886.2 to 7730.2] | 16761 [16761 to 16761]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 2903.8 [2420.8 to 6799.9] | 22000 [22000 to 22000] | 4254.2 [2074 to 8559.2] | 4811.6 [2823.2 to 13714.5] | 4119.8 [1673.6 to 8207.9] | 6705 [4218 to 8600.6] | 3609.4 [1900.9 to 12713.1]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 2903.8 [2420.8 to 6799.9] | 22000 [22000 to 22000] | 7544.4 [4787.2 to 9652.3] | 4610 [2910 to 13500.2] | 9226 [402.8 to 15873.3] | 6207.5 [3321.6 to 8959] | 3503.5 [1849.2 to 12111.9]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 24 | 24 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 3074.5 [1752.8 to 6132] | 5450.2 [3614.9 to 7521.1] | 3757.2 [1824.5 to 7062] | 4377.2 [1549.8 to 7839.9] | 5785.1 [3959.2 to 8580.8] | 8264.2 [5681.2 to 10629.8] | 6218.5 [3751 to 13401.8]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 50 | 48 | 49 | 99
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 2129 [351.1 to 4434.1] | 2121.8 [12.1 to 5765.6] | 3877.5 [2449.8 to 6245] | 4657 [2207.6 to 8233.1] | 7018.5 [3255.6 to 11673.8] | 7882 [4650.5 to 10555.5] | 4350 [2516.2 to 10204.6]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 741.8 [310.8 to 2310.2] | 1220.1 [12.1 to 4265.7] | 3970.1 [2488.4 to 5625.9] | 4713.8 [2569.2 to 8528.8] | 9034.8 [3255.6 to 13397.9] | 6215.9 [4113.8 to 9481.1] | 3454 [1593.5 to 5449.5]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru |  |  | 547.8 [153.2 to 958] | 5159.2 [2580.1 to 7608.6] | 1699.2 [1082 to 2201.1] | 1634.8 [1171.1 to 2098.4] | 3405.5 [3405.5 to 3405.5]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 2345.2 [1799.2 to 2365.4] | 4631.5 [4631.5 to 4631.5] | 1728.5 [345.2 to 2753] | 2320.2 [946.4 to 4908.1] | 1891 [1042.1 to 2935.9] | 2551.6 [2437 to 3225.2] | 1573.1 [283.2 to 2905.6]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 2345.2 [1799.2 to 2365.4] | 4631.5 [4631.5 to 4631.5] | 2346.6 [1622.2 to 3395.2] | 2211 [946.8 to 4139.2] | 3902.8 [1159.2 to 4859.9] | 2993.8 [2506.5 to 3776] | 1415.2 [189.4 to 2565]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 23 | 24 | 25 | 50
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 1367.2 [411 to 2780.2] | 4262.8 [3097.8 to 7194] | 2059.8 [310 to 6002.8] | 3125.8 [806.8 to 9861.4] | 7868.5 [3332.9 to 9858.1] | 9611.8 [5616.5 to 12570] | 3746.2 [1709.6 to 9411.6]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 49 | 48 | 49 | 99
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 488.8 [9.2 to 2020.1] | 91.2 [1 to 2734.8] | 2059.8 [562.8 to 5227.5] | 3125.8 [913.5 to 9593.2] | 7271.1 [2195.8 to 11250.9] | 7521.5 [3017.8 to 11929.5] | 2698.2 [520.1 to 7149]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 24 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 19.8 [2.2 to 568.5] | 13.4 [1 to 709.4] | 2001.6 [997.4 to 4191.4] | 2984.2 [1184.4 to 8780.8] | 6749.1 [1390.9 to 14595.4] | 4729.4 [2768.4 to 7843.6] | 630.5 [137.8 to 4620.5]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru |  |  | 175.2 [1 to 422.8] | 5091.8 [2548.1 to 6470.5] | 686.5 [246.9 to 1175.1] | 1202.9 [1052.9 to 1352.8] | 849.2 [849.2 to 849.2]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 393 [296 to 940.1] | 260.5 [260.5 to 260.5] | 243 [12.5 to 999] | 1788.8 [408.7 to 3230.5] | 747.5 [246.9 to 1774.1] | 1269.1 [1029.6 to 1497.4] | 130.9 [2.8 to 1055]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 393 [296 to 940.1] | 260.5 [260.5 to 260.5] | 721.6 [127.1 to 1071.1] | 1470.5 [466.4 to 2808.1] | 1845.2 [391.3 to 3901.2] | 1269.1 [1047.7 to 1539.4] | 126.8 [2.8 to 949.4]

5. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (BAMA IgA) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  2019-nCoV S/293F-50 at Month 0-Peru | 22 | 3 | 23 | 23 | 22 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  2019-nCoV S/293F-50 at Month 0-Total | 38 | 13 | 49 | 48 | 42 | 47 | 92
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-USA | 16 | 10 | 26 | 25 | 20 | 22 | 43
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Peru | 0 | 0 | 9 | 2 | 14 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  2019-nCoV S/293F-50 at Month 2-Total | 3 | 1 | 23 | 17 | 19 | 6 | 17
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  2019-nCoV S/293F-50 at Month 2-USA | 3 | 1 | 14 | 15 | 5 | 4 | 16
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 DB His-50 at Month 0-Peru | 18 | 3 | 21 | 21 | 22 | 25 | 47
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 DB His-50 at Month 0-Total | 27 | 12 | 38 | 41 | 40 | 45 | 80
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 DB His-50 at Month 0-USA | 9 | 9 | 17 | 20 | 18 | 20 | 33
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 DB His-50 at Month 2-Peru | 0 | 0 | 6 | 2 | 12 | 2 | 1
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 DB His-50 at Month 2-Total | 2 | 1 | 15 | 14 | 17 | 5 | 11
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 DB His-50 at Month 2-USA | 2 | 1 | 9 | 12 | 5 | 3 | 10
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 23 | 3 | 23 | 23 | 24 | 25 | 43
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 39 | 15 | 47 | 47 | 45 | 47 | 82
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 16 | 12 | 24 | 24 | 21 | 22 | 39
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 0 | 0 | 9 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 2 | 1 | 21 | 16 | 20 | 5 | 14
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 2 | 1 | 12 | 13 | 5 | 3 | 13
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 23 | 3 | 23 | 23 | 22 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 39 | 13 | 50 | 48 | 42 | 47 | 94
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 16 | 10 | 27 | 25 | 20 | 22 | 44
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 0 | 0 | 11 | 2 | 14 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 3 | 1 | 26 | 17 | 19 | 6 | 16
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 3 | 1 | 15 | 15 | 5 | 4 | 15
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 23 | 3 | 22 | 22 | 22 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 36 | 13 | 48 | 46 | 42 | 47 | 90
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 13 | 10 | 26 | 24 | 20 | 22 | 41
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 0 | 0 | 8 | 2 | 14 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 3 | 1 | 20 | 17 | 19 | 6 | 15
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 3 | 1 | 12 | 15 | 5 | 4 | 14
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 4 | 1 | 12 | 16 | 19 | 20 | 35
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 7 | 4 | 15 | 29 | 32 | 33 | 48
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 3 | 3 | 3 | 13 | 13 | 13 | 13
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 0 | 0 | 2 | 1 | 5 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 0 | 1 | 4 | 9 | 9 | 2 | 6
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 0 | 1 | 2 | 8 | 4 | 0 | 5
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 22 | 3 | 21 | 22 | 22 | 25 | 48
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 36 | 13 | 44 | 45 | 41 | 47 | 89
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 14 | 10 | 23 | 23 | 19 | 22 | 41
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 0 | 0 | 6 | 2 | 13 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 3 | 1 | 19 | 16 | 18 | 6 | 16
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 3 | 1 | 13 | 14 | 5 | 4 | 15
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 20 | 3 | 11 | 23 | 15 | 21 | 47
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 15 | 2 | 8 | 20 | 14 | 21 | 44
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 42 | 20 | 18 | 36 | 32 | 42 | 85
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 22 | 7 | 13 | 29 | 27 | 38 | 71
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 22 | 17 | 7 | 13 | 17 | 21 | 38
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 7 | 5 | 5 | 9 | 13 | 17 | 27
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 0 | 0 | 5 | 2 | 13 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 1 | 0 | 16 | 12 | 18 | 4 | 9
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 1 | 0 | 11 | 10 | 5 | 2 | 8

6. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (BAMA IgA) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
MFI
  2019-nCoV S/293F-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  2019-nCoV S/293F-250 at Month 0-Peru | 1386.2 [588 to 3401.8] | 1661.2 [1043.5 to 3932.1] | 2782.8 [1240 to 6458] | 3824.5 [2088 to 7100.5] | 8149.6 [3577 to 11434.5] | 9913.8 [5485 to 16653.5] | 3818.9 [2128.9 to 7245.1]
  2019-nCoV S/293F-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  2019-nCoV S/293F-250 at Month 0-Total | 732 [214.1 to 1944.8] | 517.5 [33.6 to 2436.8] | 1493 [701.8 to 3198] | 2831 [1075 to 6386.8] | 3937.5 [2108.6 to 8818] | 3256.9 [2269.5 to 9825.4] | 2177.2 [703.6 to 5355.9]
  2019-nCoV S/293F-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  2019-nCoV S/293F-250 at Month 0-USA | 518.8 [37 to 1083.8] | 361.2 [33.6 to 2436.8] | 999.9 [600.4 to 1651] | 1868.4 [850.3 to 5626.9] | 2831.6 [890.1 to 4766.2] | 2407.5 [1336.8 to 3196.2] | 1292.8 [390.8 to 2564.8]
  2019-nCoV S/293F-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  2019-nCoV S/293F-250 at Month 2-Peru |  |  | 457.2 [117.2 to 646.8] | 1272.2 [663.4 to 2134.2] | 2037.5 [1378.2 to 3073.2] | 4681.6 [4323.3 to 5039.9] | 8920.8 [8920.8 to 8920.8]
  2019-nCoV S/293F-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  2019-nCoV S/293F-250 at Month 2-Total | 1902.2 [1230 to 3130.4] | 4086.5 [4086.5 to 4086.5] | 642.8 [277.2 to 875.5] | 2688.1 [831.2 to 3771.1] | 1765 [397.8 to 2616.5] | 1630.2 [1159.2 to 3438.9] | 465 [361.5 to 1775.8]
  2019-nCoV S/293F-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  2019-nCoV S/293F-250 at Month 2-USA | 1902.2 [1230 to 3130.4] | 4086.5 [4086.5 to 4086.5] | 712 [519.7 to 916.8] | 2761.2 [917 to 4261.1] | 1148.9 [78.1 to 2202.4] | 1239.4 [1014.1 to 1515] | 460.8 [360.8 to 1166.5]
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  2019-nCoV S/293F-50 at Month 0-Peru | 4666 [2600.2 to 10206.8] | 6144.8 [4454.9 to 10284.4] | 8446.2 [4770 to 16894.5] | 9177.5 [5253.2 to 18415.2] | 17476.5 [11429.7 to 22000] | 22000 [14734 to 22000] | 11884.5 [6291.9 to 16184.8]
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  2019-nCoV S/293F-50 at Month 0-Total | 3158.5 [853.7 to 7593] | 2428 [139.2 to 7828.9] | 5461.2 [2735.8 to 10318.2] | 8326.5 [3622.2 to 15899.6] | 11991.2 [5031.8 to 18433.8] | 9468.2 [6621.1 to 22000] | 7086 [2970.6 to 13692.4]
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  2019-nCoV S/293F-50 at Month 0-USA | 1962.8 [184 to 3639.8] | 1705.6 [139.2 to 7828.9] | 3735.2 [2226.3 to 6124.2] | 6235.1 [2679.1 to 11670.9] | 8299.6 [3850.7 to 12724.4] | 7566.8 [4263.2 to 8878.8] | 4570 [1625.2 to 8088]
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  2019-nCoV S/293F-50 at Month 2-Peru |  |  | 1324.5 [449.5 to 2601.8] | 3951.5 [2089.6 to 6816.8] | 6588 [4829.2 to 8250.1] | 12474.9 [12384.4 to 12565.3] | 19584.8 [19584.8 to 19584.8]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  2019-nCoV S/293F-50 at Month 2-Total | 6468.8 [4381.6 to 9069.8] | 11144 [11144 to 11144] | 2494.2 [1072.2 to 3137] | 6919.2 [3324.1 to 9006.8] | 6300 [1769.1 to 7385.5] | 5126.8 [3915.5 to 10686.9] | 2111.5 [1495.4 to 4591.9]
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  2019-nCoV S/293F-50 at Month 2-USA | 6468.8 [4381.6 to 9069.8] | 11144 [11144 to 11144] | 2749.2 [2013 to 3516.9] | 6952.2 [3493.5 to 8426.4] | 4303.1 [217 to 7231.9] | 4073 [3688 to 4757.4] | 2093.5 [1463.5 to 3573.9]
  229E-RBD-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  229E-RBD-250 at Month 0-Peru | 125.2 [89.8 to 244.2] | 450 [251.6 to 697.9] | 119.2 [75.8 to 178] | 194.5 [83.8 to 320] | 161.5 [109.3 to 220.4] | 308.8 [209.5 to 491] | 175.6 [99.2 to 277.9]
  229E-RBD-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  229E-RBD-250 at Month 0-Total | 94.9 [72.6 to 158.2] | 145 [83.2 to 276.5] | 94.5 [43.8 to 169] | 177 [89.2 to 337.2] | 152.4 [99.8 to 235.9] | 236.2 [112.7 to 451.1] | 132.5 [67.5 to 252.2]
  229E-RBD-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  229E-RBD-250 at Month 0-USA | 82.2 [55.2 to 121.5] | 134.8 [79.1 to 184.4] | 76 [33.1 to 124.6] | 159.6 [104 to 353.1] | 139 [96.4 to 235.9] | 119.8 [76.2 to 247.5] | 103.2 [60.8 to 242.5]
  229E-RBD-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  229E-RBD-250 at Month 2-Peru |  |  | 68.8 [25.8 to 97] | 179 [117.8 to 197.1] | 75.5 [52.9 to 91.2] | 346.2 [278 to 414.5] | 113.2 [113.2 to 113.2]
  229E-RBD-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  229E-RBD-250 at Month 2-Total | 83 [62.9 to 84.2] | 105 [105 to 105] | 66.2 [28 to 97] | 143.2 [108.1 to 234.2] | 90.8 [68.9 to 177.5] | 258.1 [154.8 to 328.8] | 99.8 [57.7 to 179.1]
  229E-RBD-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  229E-RBD-250 at Month 2-USA | 83 [62.9 to 84.2] | 105 [105 to 105] | 66.1 [41.9 to 117] | 135 [109.1 to 264.8] | 177.5 [136.3 to 669.8] | 221.5 [115.1 to 313.9] | 99.5 [56.9 to 186.1]
  229E-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  229E-RBD-50 at Month 0-Peru | 481.5 [359 to 974.8] | 2143 [971.4 to 3283.1] | 487 [344 to 785] | 772.2 [347.2 to 983] | 599.9 [407.9 to 840.6] | 1119.2 [796.8 to 1808.8] | 654.9 [380 to 1075.3]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  229E-RBD-50 at Month 0-Total | 414.6 [267.4 to 620.8] | 595.2 [356.2 to 1040.5] | 417 [205.5 to 644.8] | 678.8 [352.1 to 1130.4] | 598 [376.7 to 822.5] | 831.2 [461.3 to 1628] | 504 [279.2 to 1013]
  229E-RBD-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  229E-RBD-50 at Month 0-USA | 340.5 [240.8 to 520.5] | 495.1 [333.2 to 869.4] | 297.5 [154.6 to 516] | 643.5 [367.3 to 1172.5] | 464.9 [336.6 to 799.4] | 476 [288.8 to 925] | 409.5 [225.8 to 984.8]
  229E-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  229E-RBD-50 at Month 2-Peru |  |  | 321 [124.8 to 388.8] | 700 [425.9 to 756] | 295.8 [204.8 to 323.1] | 1148.2 [891.9 to 1404.6] | 268.2 [268.2 to 268.2]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  229E-RBD-50 at Month 2-Total | 299.2 [224.5 to 332.9] | 382.2 [382.2 to 382.2] | 282.8 [124.8 to 388.8] | 527.9 [365.5 to 885.3] | 332.5 [234.8 to 699.9] | 786.8 [540.4 to 1137.9] | 362.6 [205.9 to 662.8]
  229E-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  229E-RBD-50 at Month 2-USA | 299.2 [224.5 to 332.9] | 382.2 [382.2 to 382.2] | 260.4 [135.6 to 430.4] | 518.8 [371.2 to 972.2] | 699.9 [447.5 to 1730.8] | 723.4 [434.7 to 1004.6] | 445 [202.5 to 687.4]
  HCoV-229E S1S2 ECD His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-229E S1S2 ECD His-250 at Month 0-Peru | 130 [101.2 to 370.5] | 328.1 [160.4 to 552.9] | 157.2 [83.5 to 221.5] | 147 [74 to 290] | 104.6 [52.1 to 253.6] | 157.5 [83.5 to 258.8] | 129.1 [66.1 to 264.1]
  HCoV-229E S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-229E S1S2 ECD His-250 at Month 0-Total | 115.1 [69.8 to 251.8] | 121.1 [80.6 to 219.2] | 86.8 [30 to 191] | 128.5 [62.9 to 285.8] | 105.9 [58.8 to 222.3] | 126.5 [66.9 to 236] | 106.8 [47 to 236.8]
  HCoV-229E S1S2 ECD His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-229E S1S2 ECD His-250 at Month 0-USA | 109.2 [34.5 to 194] | 103.5 [78.9 to 204.6] | 43.8 [18.3 to 109.8] | 104.8 [49.8 to 229.1] | 105.9 [66.8 to 205.4] | 116.8 [41 to 227] | 83.8 [30.8 to 208.5]
  HCoV-229E S1S2 ECD His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-229E S1S2 ECD His-250 at Month 2-Peru |  |  | 194.5 [102.8 to 252.5] | 238.2 [172.5 to 343.5] | 128 [66.9 to 170.1] | 379.5 [268.1 to 490.9] | 17 [17 to 17]
  HCoV-229E S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-229E S1S2 ECD His-250 at Month 2-Total | 65.2 [46.4 to 141.9] | 126.2 [126.2 to 126.2] | 109 [43 to 224] | 163.8 [85.5 to 315.5] | 166.5 [70.4 to 359.5] | 135.9 [93.6 to 271.3] | 99.1 [40.7 to 314.6]
  HCoV-229E S1S2 ECD His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-229E S1S2 ECD His-250 at Month 2-USA | 65.2 [46.4 to 141.9] | 126.2 [126.2 to 126.2] | 71.9 [39.5 to 155] | 137 [75.6 to 284.9] | 359.5 [253.1 to 460.4] | 100.8 [70.7 to 163.6] | 111.8 [44.2 to 333.4]
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-229E S1S2 ECD His-50 at Month 0-Peru | 579.2 [346.5 to 1431.8] | 1333 [715.9 to 2160.4] | 593.5 [315.5 to 954.5] | 656.2 [299.5 to 1341.5] | 440.1 [217.8 to 1022.3] | 659.2 [384 to 1027.5] | 480.1 [238.1 to 1053.6]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 487.2 [276.8 to 998.8] | 548.1 [334.9 to 975.6] | 329 [123.2 to 743.5] | 552.8 [290.1 to 1066.2] | 424.2 [243.6 to 912.2] | 542.1 [241.3 to 1008.4] | 420 [183.8 to 1053.2]
  HCoV-229E S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-229E S1S2 ECD His-50 at Month 0-USA | 465.5 [135.2 to 849] | 493 [302.9 to 901.8] | 178.4 [94.3 to 459.4] | 445.6 [234.7 to 822] | 421.5 [282.6 to 878.1] | 466.8 [162.5 to 931.5] | 364.8 [119.8 to 906]
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-229E S1S2 ECD His-50 at Month 2-Peru |  |  | 698 [374.8 to 1095] | 843.5 [562.9 to 1271.6] | 387 [212.5 to 699.5] | 1399.4 [941.2 to 1857.6] | 82.8 [82.8 to 82.8]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 278.2 [177.8 to 619] | 448.8 [448.8 to 448.8] | 447 [160.2 to 918.5] | 642.4 [285.2 to 1201.1] | 685.8 [239 to 1155] | 418.1 [314.8 to 1002.4] | 405.2 [153.7 to 976.7]
  HCoV-229E S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-229E S1S2 ECD His-50 at Month 2-USA | 278.2 [177.8 to 619] | 448.8 [448.8 to 448.8] | 273.5 [135.5 to 654.8] | 614.2 [276.8 to 1026.4] | 1155 [885.2 to 1664] | 327.6 [248.9 to 558.8] | 482.8 [162.5 to 1067.9]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Peru | 149 [114 to 192] | 124.8 [98.9 to 899.9] | 200.8 [81.8 to 380.8] | 598 [253 to 897] | 357.8 [217.4 to 988.1] | 599.2 [329.5 to 1111.2] | 289.4 [180.2 to 945.1]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Total | 153.9 [111.4 to 312.6] | 328.8 [142.2 to 1374.1] | 200.8 [82.5 to 380.8] | 680.8 [268 to 1413.8] | 483.6 [241.3 to 1503] | 634.6 [339.8 to 1276.1] | 304.8 [139 to 777.8]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-USA | 194.5 [109.8 to 354.5] | 448.6 [208.6 to 1374.1] | 186.9 [106.4 to 379.6] | 744.2 [316 to 2270.9] | 650.2 [271 to 2067.2] | 875.8 [370.8 to 1435] | 319.2 [115 to 686.2]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Peru |  |  | 142 [88 to 309.5] | 135.5 [98.6 to 351.4] | 342.8 [162.6 to 872.5] | 540.2 [485 to 595.5] | 2519 [2519 to 2519]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Total | 663 [484.9 to 983.2] | 242.8 [242.8 to 242.8] | 210.2 [134.2 to 484.5] | 749 [375.6 to 1974.3] | 379.8 [162.6 to 897.4] | 400.6 [302.1 to 595.5] | 269.1 [120.4 to 1054]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-USA | 663 [484.9 to 983.2] | 242.8 [242.8 to 242.8] | 240.2 [176.5 to 539.6] | 1333.8 [392.6 to 2461.4] | 530.9 [207.3 to 1055.9] | 325.2 [272.9 to 850.1] | 254 [116.2 to 878]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Peru | 620.8 [490.2 to 765.2] | 583.6 [488.8 to 2825.3] | 802.5 [335.8 to 1463] | 2467 [1054.8 to 3207.8] | 1471.4 [969.4 to 4263.3] | 2385.5 [1418.5 to 4160.8] | 1273.9 [704.9 to 2929.7]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 656.5 [500.4 to 1360] | 1423.4 [644.2 to 4740.1] | 802.5 [389.8 to 1556.8] | 2643.2 [1129.2 to 4805.4] | 1848.1 [1018.6 to 5324.2] | 2405.5 [1392.2 to 4271.4] | 1280.8 [568 to 2663.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-USA | 809.2 [530 to 1496.5] | 1936.9 [865.7 to 4740.1] | 882.1 [467.4 to 1597.8] | 2800.2 [1232.7 to 6306.3] | 2481.6 [1100.4 to 6433.5] | 3168.5 [1383.5 to 4673.8] | 1310 [467.8 to 2440.5]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Peru |  |  | 649.5 [280 to 1220.5] | 405 [345.4 to 1146.6] | 1766.2 [530 to 3200.4] | 1904.2 [1518.1 to 2290.4] | 6969 [6969 to 6969]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 2649.2 [1952.2 to 3733] | 947 [947 to 947] | 844.8 [459.5 to 1714.2] | 2519.5 [1349.1 to 5729.1] | 1766.2 [602.4 to 3365.8] | 1364.4 [1165.6 to 2372.9] | 1057.4 [513.4 to 3326.6]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-USA | 2649.2 [1952.2 to 3733] | 947 [947 to 947] | 933.6 [647.6 to 1851.3] | 4018.8 [1544.8 to 7106.6] | 1723.5 [842.8 to 3663.9] | 1364.4 [1161.8 to 2458] | 888.2 [493.6 to 2804.2]
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Peru | 16 [10.5 to 36.8] | 15.8 [8.9 to 22.6] | 19 [9.5 to 30.5] | 21.2 [7.2 to 37.2] | 24.5 [7.8 to 38.6] | 15.5 [1 to 38.2] | 19.6 [8.4 to 45.2]
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Total | 16.1 [10.1 to 42] | 25.9 [12.7 to 58.6] | 12.5 [6 to 26.8] | 18 [7.4 to 43.8] | 31.6 [15.3 to 59.9] | 29.1 [5.4 to 55.1] | 19.8 [8.9 to 38.1]
  HCoV-NL63 S1S2 ECD His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-NL63 S1S2 ECD His-250 at Month 0-USA | 24.5 [9.5 to 49.5] | 32.9 [16.7 to 66.6] | 9.2 [3.7 to 20.1] | 16.4 [7.7 to 44.6] | 51.6 [23.4 to 67.3] | 39.5 [24.2 to 79] | 19.8 [9.5 to 37.5]
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Peru |  |  | 15.5 [10 to 50.5] | 18.5 [11.8 to 23.8] | 16 [8.6 to 20.5] | 98 [62.5 to 133.5] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Total | 26.2 [23.1 to 43.2] | 6.2 [6.2 to 6.2] | 20.8 [8.8 to 38.2] | 18.4 [9.8 to 39.5] | 18.2 [11.2 to 49.4] | 25.2 [12.4 to 37.5] | 36.4 [18.2 to 57.8]
  HCoV-NL63 S1S2 ECD His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-NL63 S1S2 ECD His-250 at Month 2-USA | 26.2 [23.1 to 43.2] | 6.2 [6.2 to 6.2] | 21.9 [8.3 to 32.4] | 18.2 [10.5 to 41.1] | 49.4 [37.7 to 104.3] | 16.1 [6.8 to 27.9] | 39.5 [21.9 to 64]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Peru | 58 [38.8 to 134.8] | 71.9 [43.2 to 101.1] | 78.2 [41.8 to 167] | 61.2 [30 to 166.5] | 88.9 [26.6 to 153] | 21.8 [1 to 150.2] | 70.5 [33.1 to 220.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 73 [25.8 to 184.9] | 106.4 [56.1 to 208.1] | 65.2 [28.5 to 115.8] | 67.2 [30 to 173.6] | 133.4 [60 to 230.2] | 123.9 [14.6 to 221.2] | 81.8 [34.1 to 174.4]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-NL63 S1S2 ECD His-50 at Month 0-USA | 96.2 [23 to 219.5] | 150.8 [72.8 to 279.4] | 41.6 [20.7 to 108.2] | 72 [23 to 183.2] | 198.4 [99.2 to 313.1] | 186 [70.8 to 305.8] | 90.2 [36 to 145.5]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Peru |  |  | 74.2 [38 to 189] | 82 [45.4 to 85.5] | 67.2 [38.4 to 89.2] | 594.2 [444 to 744.5] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 22 | 6 | 19
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 147.5 [119.8 to 199.4] | 36.5 [36.5 to 36.5] | 81.8 [32.5 to 165.2] | 80 [37.1 to 152.1] | 87.2 [50 to 156.6] | 99.2 [26.6 to 252.9] | 98 [64.6 to 222]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 7 | 4 | 18
  HCoV-NL63 S1S2 ECD His-50 at Month 2-USA | 147.5 [119.8 to 199.4] | 36.5 [36.5 to 36.5] | 92.6 [21.2 to 147.8] | 78 [38.6 to 171.6] | 163.5 [128.6 to 455.4] | 40.5 [9.8 to 83.8] | 122.4 [79.9 to 222]
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Peru | 421.8 [305.8 to 619] | 571.1 [262.7 to 2215.8] | 621.2 [278.2 to 1361] | 1187.5 [456.5 to 1905.2] | 989.1 [345.4 to 1559] | 1213.2 [623.2 to 2450.8] | 591.9 [356.3 to 1670.1]
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Total | 481.6 [322.9 to 797.3] | 884.2 [425.2 to 2295.5] | 541 [233.8 to 1199.2] | 1386.2 [518.5 to 3339.2] | 1181 [478.1 to 2433.1] | 1302.4 [608.6 to 2482.6] | 735.8 [306.2 to 1776.8]
  HCoV-OC43 S1S2 ECD His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-OC43 S1S2 ECD His-250 at Month 0-USA | 504.5 [353.2 to 1403.5] | 954 [600.9 to 2295.5] | 509.1 [229.8 to 852.9] | 2208 [619.8 to 4864.6] | 1362.6 [603.7 to 4023.8] | 1391.5 [603.8 to 2605.8] | 772.2 [215.2 to 1808.5]
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Peru |  |  | 346 [210.5 to 993.5] | 220.8 [164.5 to 726] | 717 [282.9 to 1365.6] | 805.1 [759.1 to 851.2] | 4030.2 [4030.2 to 4030.2]
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Total | 832.8 [736.9 to 1024.4] | 612.2 [612.2 to 612.2] | 606.5 [288.5 to 1015.2] | 1748.9 [392.1 to 5996.4] | 921 [348.5 to 1765.2] | 583.2 [450.7 to 851.2] | 1088.1 [278.6 to 3229.7]
  HCoV-OC43 S1S2 ECD His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-OC43 S1S2 ECD His-250 at Month 2-USA | 832.8 [736.9 to 1024.4] | 612.2 [612.2 to 612.2] | 700.9 [295.6 to 1045.2] | 2575.5 [561.5 to 6913.4] | 1412.8 [849.5 to 1937.1] | 451.6 [432.9 to 653.8] | 1055.2 [276.6 to 2821.6]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Peru | 1669.2 [1243.5 to 2515] | 2364.9 [1164.8 to 6805.2] | 2410.2 [1124.5 to 4152.5] | 4462.8 [1807.8 to 6591.2] | 3525.2 [1489.9 to 6133.6] | 5101.8 [2537.5 to 7638.5] | 2568.4 [1635.9 to 4584.1]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 2032.4 [1340.1 to 2943.3] | 3540 [1821.3 to 8140.1] | 2171.5 [1044.2 to 4024.5] | 5032.2 [2204.9 to 8806] | 4103.4 [1941.1 to 8606.4] | 5020.8 [2513.9 to 7627.4] | 2708.8 [1175.9 to 5926.9]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  HCoV-OC43 S1S2 ECD His-50 at Month 0-USA | 2120.5 [1627 to 5052.2] | 3772.1 [2476.2 to 8140.1] | 1986.2 [983.3 to 3146.6] | 7532.8 [2586.9 to 11554.1] | 5224.1 [2340.1 to 9621.4] | 4939.8 [2506 to 7594] | 3052.8 [1043.8 to 6111.5]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Peru |  |  | 1234.2 [1066.5 to 3223.5] | 639.5 [519.1 to 2434.5] | 1990 [870.6 to 5109.4] | 2501.9 [2137.8 to 2865.9] | 9763 [9763 to 9763]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 3461.5 [2964.2 to 3968.6] | 2148 [2148 to 2148] | 2316.8 [1071.2 to 3237] | 5426.5 [1512.4 to 14248.9] | 3481 [1041.5 to 5940.8] | 1759.1 [1720.3 to 2865.9] | 4846.5 [1150.4 to 7468.7]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HCoV-OC43 S1S2 ECD His-50 at Month 2-USA | 3461.5 [2964.2 to 3968.6] | 2148 [2148 to 2148] | 2475.2 [1325.9 to 3286.7] | 7931.2 [2113.1 to 15247.9] | 4800.1 [2334.5 to 6707.9] | 1728.4 [1614.9 to 2384.9] | 3977.8 [1141.2 to 7037.5]
  HKU1-RBD-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HKU1-RBD-250 at Month 0-Peru | 97.5 [60.8 to 148.8] | 208.1 [163.2 to 310.8] | 99 [62 to 125.2] | 113.2 [75.5 to 186.5] | 169 [121.8 to 497.1] | 223.5 [136.5 to 356.2] | 134.4 [79.7 to 231.9]
  HKU1-RBD-250 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 51 | 48 | 50 | 99
  HKU1-RBD-250 at Month 0-Total | 94.9 [60.8 to 140.8] | 120.5 [65.8 to 518] | 64.2 [44 to 125.2] | 150.5 [91.8 to 221.1] | 156.9 [105.5 to 299] | 160.5 [106.8 to 317.2] | 130 [57.9 to 231.1]
  HKU1-RBD-250 at Month 0-USA: number analyzed (Participants) | 25 | 17 | 28 | 26 | 24 | 25 | 49
  HKU1-RBD-250 at Month 0-USA | 89 [61.8 to 136.5] | 115.2 [49.5 to 518] | 54 [35.8 to 108.4] | 186.4 [106.8 to 320.2] | 135.5 [85.1 to 237.8] | 116.5 [86.8 to 173.8] | 98.2 [49 to 214.2]
  HKU1-RBD-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HKU1-RBD-250 at Month 2-Peru |  |  | 52.8 [27.5 to 87.2] | 112.8 [96 to 158.2] | 95.2 [73.2 to 340.6] | 244.5 [222 to 267] | 157.2 [157.2 to 157.2]
  HKU1-RBD-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HKU1-RBD-250 at Month 2-Total | 92 [85.1 to 681.6] | 83.2 [83.2 to 83.2] | 53.2 [34.8 to 110] | 155.6 [102.4 to 246.8] | 112.5 [80.2 to 292] | 204.8 [108.8 to 269.6] | 122.9 [53.6 to 162.4]
  HKU1-RBD-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HKU1-RBD-250 at Month 2-USA | 92 [85.1 to 681.6] | 83.2 [83.2 to 83.2] | 55.1 [41.5 to 131.4] | 157.5 [106.6 to 292.4] | 132.9 [101.5 to 266.9] | 144.2 [74.7 to 268] | 108.8 [51.4 to 166.9]
  HKU1-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  HKU1-RBD-50 at Month 0-Peru | 410.5 [258.8 to 598.2] | 815.9 [628.9 to 1468] | 337.2 [273.5 to 515.2] | 410.8 [313 to 582] | 629 [476.5 to 2169] | 771.2 [508.5 to 1253] | 527 [349.7 to 845.6]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 21 | 53 | 51 | 48 | 50 | 99
  HKU1-RBD-50 at Month 0-Total | 375.9 [268.2 to 582.1] | 514.2 [301.8 to 1740.8] | 311 [185.5 to 515.2] | 568 [355.1 to 847.5] | 555 [396.2 to 1160.1] | 559.2 [374.8 to 1105.2] | 447.2 [237.8 to 862]
  HKU1-RBD-50 at Month 0-USA: number analyzed (Participants) | 25 | 17 | 28 | 26 | 24 | 25 | 49
  HKU1-RBD-50 at Month 0-USA | 373.5 [291 to 577] | 453 [233 to 1740.8] | 243.6 [147.4 to 449.6] | 686.2 [420.2 to 1316.8] | 452.9 [370.1 to 917.4] | 395.8 [308 to 673.5] | 333.5 [186.2 to 884.5]
  HKU1-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  HKU1-RBD-50 at Month 2-Peru |  |  | 172.8 [150.8 to 355] | 491.2 [373.2 to 610.2] | 364.8 [321.2 to 1068.6] | 735 [715.2 to 754.8] | 376.2 [376.2 to 376.2]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  HKU1-RBD-50 at Month 2-Total | 432.2 [362.9 to 2247.5] | 324.2 [324.2 to 324.2] | 236 [150.8 to 448.5] | 549 [403.6 to 834.7] | 397.5 [341.5 to 1051.5] | 731.5 [392.5 to 772.8] | 424.6 [201.3 to 732.5]
  HKU1-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  HKU1-RBD-50 at Month 2-USA | 432.2 [362.9 to 2247.5] | 324.2 [324.2 to 324.2] | 239.9 [150.9 to 500.6] | 561.8 [403.9 to 1024.5] | 510 [386.2 to 825.4] | 529.5 [267.4 to 1016.8] | 427.5 [179.1 to 748.8]
  NL63-RBD-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  NL63-RBD-250 at Month 0-Peru | 334 [210.8 to 448.2] | 481.8 [307.8 to 627.6] | 266.8 [181 to 463.2] | 276.8 [193.2 to 422] | 340.6 [254 to 708] | 399 [244.8 to 723] | 224.4 [128.8 to 313.9]
  NL63-RBD-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  NL63-RBD-250 at Month 0-Total | 262.8 [162.6 to 437.7] | 406.5 [193.8 to 688.9] | 232.5 [125.8 to 386.8] | 300 [160.1 to 505.8] | 402.8 [255.4 to 963.6] | 419.1 [215.6 to 873.1] | 285.5 [153.2 to 622.5]
  NL63-RBD-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  NL63-RBD-250 at Month 0-USA | 213.8 [140.5 to 342.5] | 406.5 [193.8 to 806.3] | 163.2 [90.4 to 321.8] | 355.8 [141.1 to 584.6] | 747.4 [256.4 to 1195.7] | 652.5 [200.2 to 1035.2] | 433.2 [169.8 to 833.5]
  NL63-RBD-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  NL63-RBD-250 at Month 2-Peru |  |  | 301.2 [159.8 to 460] | 312 [268.6 to 389.2] | 232.8 [139.9 to 395.8] | 424.6 [399.7 to 449.6] | 150.2 [150.2 to 150.2]
  NL63-RBD-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  NL63-RBD-250 at Month 2-Total | 176 [166.6 to 217.4] | 192 [192 to 192] | 180.5 [115 to 421] | 375 [227.1 to 468.9] | 332.2 [180.4 to 1064.1] | 300.8 [183.1 to 449.6] | 431.6 [261.6 to 1074.9]
  NL63-RBD-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  NL63-RBD-250 at Month 2-USA | 176 [166.6 to 217.4] | 192 [192 to 192] | 166.2 [90.8 to 289] | 405.8 [186.5 to 594.9] | 1064.1 [794.1 to 1494.8] | 197.6 [159.9 to 376.9] | 455 [319 to 1096.8]
  NL63-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  NL63-RBD-50 at Month 0-Peru | 1297.8 [898.2 to 1782] | 1837.9 [1173.8 to 2635.2] | 1098.8 [745.8 to 1894.2] | 1158.5 [806.8 to 1773.2] | 1375.9 [955.4 to 2272.4] | 1543 [912.5 to 2466.5] | 955.1 [531.1 to 1364]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  NL63-RBD-50 at Month 0-Total | 1133 [668 to 1771.5] | 1747.6 [855.1 to 3276.6] | 862 [545.2 to 1582.5] | 1160.8 [673.5 to 2169] | 1706.6 [968.9 to 3644.6] | 1683.9 [873.7 to 3427.7] | 1166.5 [588.8 to 2450.1]
  NL63-RBD-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  NL63-RBD-50 at Month 0-USA | 877.2 [638.8 to 1707.8] | 1747.6 [855.1 to 3473.1] | 659.6 [394.1 to 1305.4] | 1478 [618.4 to 2458.9] | 2868 [1116.1 to 4143.1] | 2510.8 [839.2 to 4327.2] | 1751.5 [721.8 to 3389.5]
  NL63-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  NL63-RBD-50 at Month 2-Peru |  |  | 1289.2 [648.2 to 1866.5] | 1186.8 [957 to 1565.1] | 942.5 [595.5 to 1471.5] | 1347.6 [1198.2 to 1497.1] | 423.8 [423.8 to 423.8]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  NL63-RBD-50 at Month 2-Total | 712.2 [658.1 to 873] | 774.8 [774.8 to 774.8] | 766 [439 to 1800] | 1368.5 [779.4 to 2033.7] | 1185.8 [756.1 to 3509.8] | 959.2 [739.2 to 1497.1] | 1793.6 [1094.2 to 3507.8]
  NL63-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  NL63-RBD-50 at Month 2-USA | 712.2 [658.1 to 873] | 774.8 [774.8 to 774.8] | 642 [385.8 to 1201.1] | 1467.5 [699.4 to 2217.4] | 3509.8 [2735.2 to 4470.2] | 782.8 [678.4 to 1388.8] | 1932.8 [1292.1 to 3567.5]
  OC43-RBD-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  OC43-RBD-250 at Month 0-Peru | 89 [56 to 162] | 431.6 [303.3 to 671.7] | 73.2 [59 to 150] | 103.8 [68 to 166] | 138.4 [78.4 to 254.2] | 223.2 [125.2 to 272] | 165.8 [89.6 to 230.6]
  OC43-RBD-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  OC43-RBD-250 at Month 0-Total | 108 [65.2 to 211.5] | 182.4 [101.6 to 399.7] | 73.2 [45.5 to 152.5] | 142.8 [85.6 to 254.4] | 161.9 [82.9 to 301.8] | 160.4 [81.9 to 266.4] | 108.2 [68.5 to 252.9]
  OC43-RBD-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  OC43-RBD-250 at Month 0-USA | 146.2 [67 to 248] | 163.5 [91.5 to 322.7] | 80.6 [43.8 to 217.6] | 162.9 [99.3 to 318.1] | 204 [122.9 to 330.1] | 123.2 [78 to 195.5] | 100.8 [51.5 to 282.2]
  OC43-RBD-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  OC43-RBD-250 at Month 2-Peru |  |  | 57.2 [47 to 91.5] | 123.2 [102 to 128] | 76.8 [59.4 to 148.5] | 476.6 [319.1 to 634.2] | 166.8 [166.8 to 166.8]
  OC43-RBD-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  OC43-RBD-250 at Month 2-Total | 237.5 [152.4 to 303.2] | 55.8 [55.8 to 55.8] | 83.8 [52.5 to 250.8] | 173.5 [116.7 to 335.8] | 139.8 [67 to 207.6] | 311.5 [157.9 to 497.7] | 151.2 [65.6 to 248.4]
  OC43-RBD-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  OC43-RBD-250 at Month 2-USA | 237.5 [152.4 to 303.2] | 55.8 [55.8 to 55.8] | 98.1 [71.4 to 264.9] | 239 [119.6 to 404] | 189.1 [130.9 to 223.9] | 309.1 [135.4 to 473.6] | 135.8 [59.9 to 249.4]
  OC43-RBD-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  OC43-RBD-50 at Month 0-Peru | 343.5 [233 to 566.8] | 2130.2 [1226.1 to 3186.4] | 323.5 [214 to 654.5] | 413 [270.8 to 730] | 469.9 [300.9 to 939.2] | 776.2 [396.8 to 1088.2] | 571 [332.8 to 865.6]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  OC43-RBD-50 at Month 0-Total | 472.4 [265.7 to 945.4] | 793.9 [448.9 to 1747.9] | 326.2 [193.5 to 671.8] | 524.5 [302.4 to 1055.1] | 605 [344.2 to 1110.3] | 606.8 [337.8 to 1015.2] | 431.5 [289.5 to 885.6]
  OC43-RBD-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  OC43-RBD-50 at Month 0-USA | 596.8 [322.2 to 1037.8] | 671.8 [383.1 to 1202.5] | 329.2 [190 to 836.1] | 698.2 [388.6 to 1385.8] | 786.1 [479.4 to 1173.1] | 476 [300.2 to 829] | 388 [225.2 to 1152.5]
  OC43-RBD-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  OC43-RBD-50 at Month 2-Peru |  |  | 276.8 [183 to 432.2] | 477.8 [380.8 to 597.9] | 299 [249.9 to 668] | 2104.2 [1277.8 to 2930.8] | 588 [588 to 588]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  OC43-RBD-50 at Month 2-Total | 1043.5 [644.2 to 1307.5] | 225.2 [225.2 to 225.2] | 328.2 [228.2 to 1016.8] | 745.4 [481.1 to 1251.4] | 552.2 [269.4 to 715.2] | 1226.1 [528.1 to 1982.5] | 594.4 [259.8 to 1013.1]
  OC43-RBD-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  OC43-RBD-50 at Month 2-USA | 1043.5 [644.2 to 1307.5] | 225.2 [225.2 to 225.2] | 387.6 [288.1 to 1080.4] | 914.5 [491.5 to 1575.2] | 653.8 [531.9 to 765.4] | 1226.1 [617.6 to 1790] | 600.8 [240 to 1039]
  SARS-CoV-2 DB His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 DB His-250 at Month 0-Peru | 543 [240.8 to 1479.8] | 910.1 [620.4 to 1934.7] | 1318.8 [588 to 2936] | 1897.5 [993 to 3614.8] | 3860.9 [1681.3 to 5231.6] | 4564.5 [2671 to 7601.2] | 2018.4 [909 to 4491.8]
  SARS-CoV-2 DB His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 DB His-250 at Month 0-Total | 303.1 [97.4 to 782.1] | 258.5 [45.3 to 1047.9] | 588 [256.5 to 1764.5] | 1140.5 [382.9 to 2695.8] | 1701.8 [634.2 to 4165.8] | 1595.6 [646.2 to 4467.4] | 868.8 [334.9 to 2732.9]
  SARS-CoV-2 DB His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 DB His-250 at Month 0-USA | 149.8 [35.2 to 459.8] | 180.8 [45.3 to 1040.4] | 440 [133.5 to 651.7] | 630.4 [324.4 to 1885.5] | 1050.4 [230.1 to 1778.2] | 637.8 [287 to 1144.8] | 425.8 [133.2 to 809.8]
  SARS-CoV-2 DB His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 DB His-250 at Month 2-Peru |  |  | 161.2 [58.2 to 517.2] | 617.2 [370.4 to 1068.1] | 1100.5 [695.5 to 2026.2] | 2382.8 [2142.9 to 2622.6] | 1853.8 [1853.8 to 1853.8]
  SARS-CoV-2 DB His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 DB His-250 at Month 2-Total | 280.8 [227.4 to 521.4] | 2368.8 [2368.8 to 2368.8] | 260 [99 to 517.2] | 809.8 [427.2 to 1970.7] | 994.2 [279.2 to 1886.9] | 1104 [500.2 to 1821.6] | 245.6 [126.7 to 444.1]
  SARS-CoV-2 DB His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 DB His-250 at Month 2-USA | 280.8 [227.4 to 521.4] | 2368.8 [2368.8 to 2368.8] | 290 [112.5 to 480.6] | 1002.2 [432.5 to 2279.8] | 654 [98.3 to 1554.2] | 543.6 [380.2 to 867.2] | 211.5 [125.6 to 409.6]
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 DB His-50 at Month 0-Peru | 2304.8 [767.8 to 5899.5] | 3538 [1690.7 to 7010.9] | 4670 [2052 to 8169.8] | 4758 [2425 to 8798.2] | 8992.6 [5308 to 13508.6] | 12178.5 [7477.2 to 16828] | 6193.8 [2862.4 to 12000.1]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 DB His-50 at Month 0-Total | 1250.9 [372 to 2932.6] | 1150.9 [178.3 to 4541.8] | 2052 [736.5 to 4930.2] | 3225.2 [1563.9 to 7628.8] | 5402.9 [2225.8 to 9744.4] | 5477.4 [1864.6 to 12046.4] | 2882.5 [1257.5 to 7792.4]
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 DB His-50 at Month 0-USA | 620 [151.8 to 1902] | 871.2 [152 to 3467.7] | 1672.4 [640.9 to 2139.8] | 1991.4 [1343.7 to 4912.1] | 3021.2 [849.7 to 5527.8] | 1765.2 [1092.8 to 3799] | 1591.2 [498.2 to 2882.5]
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 DB His-50 at Month 2-Peru |  |  | 692 [222.5 to 1916.8] | 1909.5 [1261.4 to 3380.4] | 3837.5 [2585 to 6053.1] | 6267.4 [5638.1 to 6896.7] | 7420.2 [7420.2 to 7420.2]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 DB His-50 at Month 2-Total | 1194.8 [912.8 to 2107.6] | 6779.5 [6779.5 to 6779.5] | 1022.2 [366.2 to 1916.8] | 2117.6 [1493.3 to 5386.8] | 3611.5 [938.2 to 5729.2] | 3749 [2084.6 to 5080.6] | 884.2 [531.9 to 2100.1]
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 DB His-50 at Month 2-USA | 1194.8 [912.8 to 2107.6] | 6779.5 [6779.5 to 6779.5] | 1055.1 [388.4 to 1864.8] | 2325.8 [1541.4 to 5556] | 2308.2 [269.8 to 5089.8] | 2219.5 [1586.8 to 3143.1] | 858.2 [504.1 to 1718.9]
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Peru | 234.8 [100.8 to 483.8] | 457.4 [336.5 to 554.4] | 506 [166 to 1150] | 1170.8 [528.5 to 4269.2] | 1406.2 [892.3 to 6171.4] | 3855.2 [2199.8 to 6346.8] | 569 [285.2 to 1947.4]
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Total | 128.9 [78.9 to 398.9] | 86.1 [55.8 to 413.8] | 335.8 [143.5 to 920.5] | 769 [221.4 to 2239.2] | 1041 [354.1 to 2154.2] | 2402 [568.1 to 5530.1] | 361.8 [125.6 to 1214]
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-USA | 84.2 [45.8 to 215] | 81.2 [55.8 to 249.2] | 253.1 [131.4 to 554.4] | 483.6 [210.8 to 1744.6] | 634.5 [174.2 to 1612.4] | 1066.2 [366.2 to 2604.2] | 239.2 [107.5 to 497.8]
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Peru |  |  | 108.2 [54.8 to 217] | 651 [383.8 to 1409.1] | 256.5 [159 to 749.6] | 1382.6 [1265.2 to 1500.1] | 303.2 [303.2 to 303.2]
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Total | 162.5 [113.5 to 762.2] | 348.8 [348.8 to 348.8] | 109.2 [68.2 to 222.8] | 344.1 [157.7 to 726.1] | 256.5 [141.1 to 836.1] | 809.5 [274 to 1500.1] | 164.4 [81.8 to 315.6]
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-USA | 162.5 [113.5 to 762.2] | 348.8 [348.8 to 348.8] | 111.2 [81.4 to 292.2] | 323.2 [163.1 to 717.4] | 265.2 [99.9 to 835.1] | 339.8 [176.9 to 967.2] | 129.5 [74.9 to 307.1]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 1028.8 [457 to 2128.2] | 2256.1 [1397.9 to 2856.5] | 2037.2 [797.5 to 4537] | 4512.5 [2344.5 to 8401.2] | 5091.6 [3741.6 to 16792] | 12226 [7813.5 to 15799.2] | 2402 [1168.5 to 6867.8]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 542.1 [318.9 to 1765.8] | 395.2 [227.8 to 1723.1] | 1603.2 [650.2 to 3705.2] | 3119.5 [910.2 to 7749.6] | 3996.6 [1441.1 to 7093.4] | 8303.8 [2277.8 to 15231.6] | 1466.8 [555.9 to 4147.4]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 357.5 [204.8 to 783.2] | 352.5 [227.8 to 1284.9] | 1095.6 [511.4 to 2274.6] | 1966 [841 to 6227.4] | 2289 [771.1 to 5483.6] | 3912.8 [1297.8 to 9189] | 1033.8 [425.8 to 1992.8]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru |  |  | 653 [278.8 to 870.2] | 2536.5 [1546.8 to 4367] | 971.2 [682.1 to 2768.1] | 3870.6 [3818.4 to 3922.8] | 1310.2 [1310.2 to 1310.2]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 713 [461.1 to 2752.8] | 1427.5 [1427.5 to 1427.5] | 434 [292.2 to 876.2] | 1435.9 [634.8 to 2686.3] | 971.2 [546.2 to 3163.5] | 3049.4 [1163.2 to 3922.8] | 684.6 [244.6 to 1340.7]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 713 [461.1 to 2752.8] | 1427.5 [1427.5 to 1427.5] | 433.1 [302 to 1145.2] | 1380 [701.8 to 2458.5] | 965.9 [271.1 to 3252.9] | 1553 [641.3 to 3857.6] | 590.8 [239.8 to 1346.4]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Peru | 510.8 [180 to 1516.8] | 812.8 [455.9 to 1843.9] | 1166.8 [350.5 to 2918.5] | 1742.2 [625.8 to 3278.5] | 3140.5 [1594 to 4530.1] | 4241.2 [2460.5 to 8315] | 1891.2 [1024.6 to 4645.2]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Total | 256.2 [84.8 to 702.6] | 218.6 [6.4 to 1063.3] | 430 [234.5 to 1174.2] | 1299 [328 to 2634.8] | 1764.9 [503.6 to 3227.9] | 1754.2 [544.5 to 4328.8] | 1069.8 [293.1 to 2767.4]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-USA | 105.8 [12.8 to 273] | 179.6 [6.4 to 928.2] | 370.5 [208.3 to 502.1] | 559.2 [276.3 to 2048.8] | 910.2 [255.4 to 1809.3] | 536 [294 to 1368.8] | 435 [124.2 to 1076]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Peru |  |  | 119.2 [56.2 to 359.5] | 556 [287.5 to 891.1] | 1057.5 [792.5 to 1489.2] | 2268.9 [2013.2 to 2524.6] | 5367.8 [5367.8 to 5367.8]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Total | 651.5 [484.1 to 875.8] | 3036 [3036 to 3036] | 238.8 [84 to 382.8] | 1083.2 [271.9 to 1416.2] | 846.5 [162.5 to 1401] | 628.9 [304.4 to 1506.1] | 176 [133.8 to 544.1]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-USA | 651.5 [484.1 to 875.8] | 3036 [3036 to 3036] | 277.6 [179.4 to 384.1] | 1146 [279.5 to 1504] | 347.9 [17.5 to 770.9] | 371.5 [237.2 to 567.3] | 169.5 [129.8 to 378.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 2082.8 [1030.2 to 5188.5] | 3215.4 [2375.1 to 5986.1] | 3899.2 [1348 to 8463] | 4311.2 [2194.8 to 8428.8] | 8338.5 [4221.9 to 11994.6] | 12204.2 [6914.2 to 16983.8] | 6274.6 [3227.6 to 10836.3]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 1067.5 [366.2 to 2900.6] | 1054.1 [35.4 to 3684.1] | 1916.8 [1067 to 4190.5] | 3689 [1292.8 to 6751.8] | 4588.2 [2000 to 8662.9] | 4657.1 [1730.1 to 12233.3] | 3352.5 [1296.4 to 8296.8]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 524.2 [43.5 to 1166] | 882.6 [28.4 to 3411.5] | 1471.2 [842.5 to 2083.1] | 2267.5 [961.9 to 4534.2] | 3400.2 [1085.6 to 5620.3] | 1804 [1160.2 to 4016.8] | 1629.2 [495.2 to 3443.8]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru |  |  | 593 [232 to 1460.2] | 1977.2 [1042.5 to 3139.4] | 3117.2 [2803.5 to 5018.5] | 6224.2 [5663.6 to 6784.9] | 14234.2 [14234.2 to 14234.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 2534.8 [2007.8 to 3078.8] | 9878 [9878 to 9878] | 988.8 [332.2 to 1574.2] | 2346.5 [1269.6 to 4247.1] | 2881.5 [742.8 to 4497.8] | 2239.6 [1177.1 to 4512.1] | 850.8 [619.5 to 1840.3]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 2534.8 [2007.8 to 3078.8] | 9878 [9878 to 9878] | 1068.1 [839.1 to 1611.7] | 2715.8 [1293.5 to 4572.1] | 1429.5 [37.9 to 2831.7] | 1364.6 [945.9 to 1989.7] | 841.2 [591.8 to 1195.8]
  SARS-CoV-2 S1 C His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1 C His-250 at Month 0-Peru | 365.8 [130.2 to 1226.8] | 507.2 [296.6 to 1384.8] | 883.5 [385 to 3011.5] | 1819.2 [791 to 3136.8] | 3305.6 [1119.6 to 5415.2] | 4220.8 [1798.5 to 8442] | 1587 [553.6 to 3450.3]
  SARS-CoV-2 S1 C His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1 C His-250 at Month 0-Total | 151.5 [32.2 to 495.8] | 117.2 [14.8 to 744.3] | 412 [152 to 977.8] | 970.5 [238.6 to 2283.6] | 1273.2 [387.6 to 3416.2] | 1327 [338.4 to 4201.5] | 644.5 [223.6 to 2004.8]
  SARS-CoV-2 S1 C His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1 C His-250 at Month 0-USA | 54.2 [4.5 to 203.2] | 106.9 [14.8 to 744.3] | 299.8 [100.4 to 430.4] | 401.2 [176.9 to 1677.7] | 612 [101.3 to 1486.4] | 334.2 [210.5 to 886.8] | 276.8 [67.5 to 665.5]
  SARS-CoV-2 S1 C His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1 C His-250 at Month 2-Peru |  |  | 90.8 [16.2 to 170.8] | 328.5 [182.4 to 651.4] | 734.2 [307.6 to 1303.2] | 1439.1 [1285.2 to 1593.1] | 1564.5 [1564.5 to 1564.5]
  SARS-CoV-2 S1 C His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1 C His-250 at Month 2-Total | 140.5 [108.1 to 323] | 639.2 [639.2 to 639.2] | 119.8 [40.2 to 261.2] | 564.4 [142.7 to 974.2] | 496.2 [121 to 1055.2] | 497.4 [282.9 to 1006.6] | 115.5 [44 to 206.4]
  SARS-CoV-2 S1 C His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1 C His-250 at Month 2-USA | 140.5 [108.1 to 323] | 639.2 [639.2 to 639.2] | 162.6 [45.9 to 278.2] | 800.2 [151.1 to 1051.8] | 288 [33.5 to 527] | 309.4 [209.3 to 429.8] | 104.2 [40 to 192.2]
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 1579.5 [367.5 to 4783.5] | 2320.9 [1088.8 to 5366.1] | 3205.2 [1713.8 to 9341] | 5855.5 [1946 to 9810.2] | 9250.4 [4361.8 to 13217.6] | 11542.8 [6017 to 17961.5] | 5657.2 [2255.9 to 10684.1]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 826.1 [163.9 to 2260.2] | 578.2 [50.9 to 3341.9] | 1713.8 [635.8 to 4561.5] | 2875.8 [928.6 to 6921.5] | 4361.5 [1375.6 to 10423.9] | 4292.2 [1470.4 to 11388.4] | 2317.8 [793.9 to 6852.5]
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 264.8 [44.5 to 902.2] | 506.1 [49.1 to 3294.1] | 1481.5 [452 to 1939.3] | 1652.4 [648.5 to 5173.1] | 2609.6 [530 to 4407.4] | 1475.5 [915.2 to 3036.5] | 1080 [328 to 2317.8]
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1 C His-50 at Month 2-Peru |  |  | 429.5 [71 to 760.5] | 1005.5 [593.5 to 2221.4] | 2455.5 [1007.6 to 4413.8] | 4198.9 [3810.4 to 4587.3] | 6491 [6491 to 6491]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 587 [464.9 to 1346.8] | 2490 [2490 to 2490] | 544 [125.5 to 1029.2] | 1655.2 [562.1 to 3330.9] | 1840.8 [469.1 to 3324.5] | 2145.2 [1365.1 to 3141.9] | 541.8 [202.8 to 791.4]
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 587 [464.9 to 1346.8] | 2490 [2490 to 2490] | 610.2 [181.5 to 1081.2] | 2212 [605.4 to 3273] | 1178.2 [101.3 to 2022.9] | 1573 [930.1 to 2067] | 519.8 [193.8 to 681.2]
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Peru | 451.5 [277.2 to 982] | 834.8 [519.5 to 1513] | 850.5 [547.8 to 1614] | 1633.8 [773.2 to 3279] | 2386.4 [1448.7 to 3207.9] | 2742.8 [1663.2 to 6081.2] | 1843.9 [1082.8 to 3064.1]
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Total | 307.8 [131.7 to 903.5] | 462.2 [175.5 to 1159.6] | 733.2 [319.8 to 1361.8] | 1427 [481.4 to 2937.4] | 1636.8 [850 to 2998.5] | 1672.2 [783.1 to 4268.8] | 1109.8 [383.2 to 2421.4]
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-USA | 189.8 [30.2 to 637.2] | 352.6 [80.6 to 1159.6] | 621.5 [251.6 to 941.8] | 1116 [469.8 to 2145.4] | 1168 [568 to 2376.1] | 1290 [394.2 to 2213.8] | 439.2 [222.8 to 1428.8]
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Peru |  |  | 346 [215.2 to 1155.5] | 900.8 [508 to 2845] | 1152 [798.8 to 1370.6] | 5372.2 [4912.4 to 5832.1] | 3516.2 [3516.2 to 3516.2]
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Total | 906.2 [685.5 to 991.2] | 1324.5 [1324.5 to 1324.5] | 709.8 [294.2 to 1155.5] | 1549.9 [685.8 to 3743.4] | 1152 [491.8 to 1459.5] | 1364.5 [825.2 to 3743.8] | 1102 [320.8 to 1512]
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-USA | 906.2 [685.5 to 991.2] | 1324.5 [1324.5 to 1324.5] | 769.1 [336.8 to 1141.8] | 1958.5 [747.2 to 3740.2] | 1008.9 [161.6 to 1693.8] | 920.6 [688.2 to 1238] | 1041.2 [311.1 to 1348.8]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 2012.8 [1248 to 3929.2] | 3682.1 [2565.7 to 5712.9] | 3802.2 [2311.5 to 6288.8] | 6633.5 [3774.8 to 11760.2] | 8764.4 [5625.3 to 11090.9] | 10069.8 [6482.2 to 17653.5] | 6459.8 [4079.4 to 9182.3]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 1355.5 [524.2 to 3653.7] | 1732.8 [624.4 to 4565.5] | 3250.2 [1414.5 to 5353.8] | 5355.2 [2139.2 to 10999.1] | 6353.6 [3592.3 to 10081.1] | 6586.8 [3121.6 to 12902.6] | 4322.5 [1640 to 7954.5]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 859.2 [147.2 to 2892.8] | 1559 [290.8 to 4565.5] | 2830.9 [1219.4 to 3997.7] | 4557.2 [2090.8 to 8041.7] | 5069.8 [2413.9 to 6825.4] | 5087.2 [1700.2 to 8646.5] | 1926 [955.8 to 5027.2]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru |  |  | 1443.8 [722.5 to 4231] | 2952 [1700.6 to 8363.9] | 4357.2 [2989.8 to 5413.9] | 12948.8 [12857.4 to 13040.1] | 9814.5 [9814.5 to 9814.5]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 3765.8 [2861.2 to 3985.6] | 4734.8 [4734.8 to 4734.8] | 2989 [1174.2 to 4159.5] | 4578.6 [2529.6 to 11753.1] | 4357.2 [2178.8 to 5596.4] | 4247.4 [3708.1 to 10668.9] | 3859.6 [1524.5 to 4881.4]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 3765.8 [2861.2 to 3985.6] | 4734.8 [4734.8 to 4734.8] | 3106 [1327.9 to 3862.1] | 4780.2 [2942.1 to 11726.4] | 3620.9 [554.1 to 6178.8] | 3844.5 [3154.2 to 4182.3] | 3751.8 [1315 to 4706.2]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Peru | 940.5 [386.5 to 2845.5] | 1380.5 [940.1 to 2492.4] | 1504.5 [656.2 to 3795.2] | 2827.2 [1783 to 4365.5] | 5367.2 [2407.3 to 7182.3] | 6622 [3348.2 to 10889] | 4030.1 [2057.6 to 6474.2]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Total | 655.8 [207.1 to 1392.2] | 483.2 [41.4 to 2353.8] | 1066.2 [426.5 to 2060.8] | 2359 [753.5 to 4325] | 3228.4 [1526.6 to 5999.6] | 3018.9 [1434.8 to 7059.8] | 2002.8 [642.4 to 5018.6]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-USA | 429.5 [48.5 to 660.5] | 363.1 [41.4 to 2353.8] | 682 [409.3 to 1345.4] | 1591.2 [534.7 to 3476.8] | 2092.8 [762.6 to 4682] | 1435.8 [762 to 2754.8] | 949.2 [350 to 2002.8]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Peru |  |  | 341.2 [114.8 to 621.2] | 983 [531.2 to 1642.9] | 1913 [1103.6 to 2892.4] | 3588.2 [3150 to 4026.5] | 12174 [12174 to 12174]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Total | 1405.5 [1058.5 to 3207.1] | 3051.2 [3051.2 to 3051.2] | 510.8 [205 to 918] | 1791.1 [710.8 to 3240.8] | 1777.5 [430.5 to 2505.9] | 2252.1 [959.1 to 3027.7] | 473.6 [340.9 to 1544.6]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-USA | 1405.5 [1058.5 to 3207.1] | 3051.2 [3051.2 to 3051.2] | 868.9 [452.7 to 955.2] | 1886.5 [812.9 to 3299.4] | 1139 [65.8 to 1802.1] | 1236.9 [663.4 to 2127.6] | 409.5 [336.6 to 1017.9]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 3373.2 [1536.2 to 7157.8] | 5532.8 [2943.7 to 9198.6] | 5187.2 [2515.5 to 11161] | 7723.8 [4711.2 to 13375] | 11580.9 [7287.9 to 17208.5] | 17681.5 [10206.2 to 22000] | 11726.9 [6183.8 to 16206.1]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 50 | 22 | 53 | 51 | 48 | 50 | 99
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 2696.9 [852.4 to 5018.1] | 2161.9 [159.9 to 9057.2] | 3981.8 [1759.2 to 6511.5] | 7053.5 [2527.9 to 11267.1] | 9034.9 [4407.8 to 14598.1] | 8970 [4342.2 to 17536.8] | 6778.2 [2671.5 to 13436.4]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 25 | 18 | 28 | 26 | 24 | 25 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 1917.2 [184 to 3080.2] | 1679 [159.9 to 9057.2] | 2949.5 [1690 to 4343.1] | 5716.9 [1983.2 to 8939.8] | 6613.6 [2719.8 to 12047.6] | 4108.2 [2701.2 to 7600] | 3418.8 [1545.5 to 6778.2]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru |  |  | 1039.8 [582.2 to 2282.8] | 3087.5 [1707 to 5127.6] | 5526.5 [3651.4 to 7994.2] | 8850.6 [7892.6 to 9808.7] | 22000 [22000 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 5119.8 [3968.1 to 8922.5] | 9059.5 [9059.5 to 9059.5] | 2231.5 [928 to 3058.8] | 5186.1 [2661.5 to 7748.6] | 5463 [1833.9 to 7410.1] | 6261.1 [3649.4 to 7180.7] | 2042.5 [1388.1 to 4885]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 5119.8 [3968.1 to 8922.5] | 9059.5 [9059.5 to 9059.5] | 2792.8 [1781 to 3846.6] | 5510.2 [2964.2 to 8096.2] | 3929.5 [183.2 to 6048.1] | 4295.5 [2871.5 to 6006.5] | 1991.5 [1382 to 3244.6]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Peru: number analyzed (Participants) | 20 | 3 | 11 | 23 | 15 | 21 | 47
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Peru | 219.4 [64 to 482.5] | 166.8 [87.5 to 232] | 248.8 [42.2 to 645.5] | 735 [185.6 to 1681.5] | 1408 [825.8 to 6131.5] | 2562 [1195 to 4096.5] | 1141.8 [401.2 to 2333.9]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Total: number analyzed (Participants) | 42 | 20 | 18 | 36 | 32 | 42 | 85
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Total | 82.9 [13.1 to 297.1] | 30.8 [6.7 to 148.8] | 144.2 [43.8 to 556.8] | 424.6 [62.1 to 1128.5] | 825.8 [148.3 to 1768.2] | 993.9 [322.2 to 2676] | 479 [119 to 1701.8]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-USA: number analyzed (Participants) | 22 | 17 | 7 | 13 | 17 | 21 | 38
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-USA | 16.8 [7.7 to 117.4] | 26.5 [5.8 to 91.8] | 69.5 [46.2 to 210.6] | 157.2 [46.5 to 410] | 275.5 [79 to 885.5] | 331 [96.2 to 629.2] | 182.9 [23.1 to 500.1]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Peru |  |  | 37.2 [11.8 to 66.8] | 165.5 [86.2 to 1830.4] | 355.2 [88.6 to 1011.6] | 1065.4 [943.6 to 1187.2] | 774.2 [774.2 to 774.2]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Total | 46.5 [46.2 to 88.5] | 43.8 [43.8 to 43.8] | 58.8 [26.8 to 84] | 248.1 [47.4 to 559.9] | 248.8 [79 to 597.2] | 164.4 [72.5 to 666.3] | 41.5 [16.1 to 226.7]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-USA | 46.5 [46.2 to 88.5] | 43.8 [43.8 to 43.8] | 62.1 [43.9 to 93.2] | 330.8 [47.8 to 557.9] | 171.9 [26.5 to 261.6] | 91.2 [51.1 to 146.6] | 38.5 [14.1 to 89]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 20 | 3 | 11 | 23 | 15 | 21 | 47
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 981 [278.1 to 2451.1] | 981.8 [517.1 to 1186.8] | 1302.2 [241.9 to 3154] | 3766.2 [791 to 6982.5] | 6168.2 [3710.9 to 16496.9] | 9308.2 [4772.2 to 14115] | 5188.8 [1739.6 to 9367]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 42 | 20 | 18 | 36 | 32 | 42 | 85
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 383.8 [65.6 to 1308.9] | 136.6 [33.3 to 701] | 680.4 [210.2 to 2929.4] | 1853.9 [310.2 to 5121.7] | 3545.8 [688.2 to 7389.3] | 3956.8 [1477.6 to 9763.5] | 2181.8 [512 to 7634.2]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 22 | 17 | 7 | 13 | 17 | 21 | 38
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 83.1 [40 to 541] | 94.2 [22.2 to 451] | 431.8 [231 to 1048.4] | 917 [213.8 to 1827.2] | 1256.2 [360.5 to 3764.8] | 1590.5 [446.5 to 2773.2] | 836.2 [123.1 to 2368.7]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 0 | 13 | 3 | 15 | 2 | 1
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru |  |  | 189 [44.8 to 435.2] | 579.8 [302.5 to 5607.9] | 1510.8 [431.6 to 3538.4] | 3434.4 [3247.3 to 3621.4] | 3687.2 [3687.2 to 3687.2]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 3 | 1 | 29 | 18 | 23 | 6 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 214.8 [212.8 to 383.6] | 176.2 [176.2 to 176.2] | 254.5 [145.5 to 435.2] | 1045.5 [219.2 to 2319.1] | 1118.8 [407.9 to 2273.8] | 776.4 [290.6 to 2512.9] | 141.9 [63.4 to 960.1]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 3 | 1 | 16 | 15 | 8 | 4 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 214.8 [212.8 to 383.6] | 176.2 [176.2 to 176.2] | 265.5 [147.9 to 398.1] | 1357.2 [220 to 2245.4] | 704.1 [64.2 to 1122.1] | 421 [158.7 to 729.1] | 139.8 [59.4 to 430.4]

7. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Enrollment Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and enrollment group among America Cohort (USA and Peru only)
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Asymptomatic, age 18 - 55
- Group 2: Asymptomatic, age 55+
- Group 3: Symptomatic, age 18 - 55
- Group 4: Symptomatic, age 55+
- Group 5: Hospitalized, age 18 - 55
- Group 6: Hospitalized, age 55+
- Group 7: Clinical spectrums
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  VRC7480_G614 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 49
  VRC7480_G614 at Month 0-Peru | 22 | 3 | 23 | 22 | 23 | 25 | 49
  VRC7480_G614 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 51 | 48 | 50 | 98
  VRC7480_G614 at Month 0-Total | 37 | 15 | 51 | 47 | 43 | 49 | 93
  VRC7480_G614 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 25 | 49
  VRC7480_G614 at Month 0-USA | 15 | 12 | 28 | 25 | 20 | 24 | 44
  VRC7480_G614 at Month 12-Peru: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 6
  VRC7480_G614 at Month 12-Peru |  |  | 1 |  |  |  | 6
  VRC7480_G614 at Month 12-Total: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 3 | 15
  VRC7480_G614 at Month 12-Total |  | 1 | 2 | 1 | 1 | 3 | 14
  VRC7480_G614 at Month 12-USA: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 3 | 9
  VRC7480_G614 at Month 12-USA |  | 1 | 1 | 1 | 1 | 3 | 8
  VRC7480_G614 at Month 2-Peru: number analyzed (Participants) | 17 | 2 | 20 | 14 | 22 | 17 | 14
  VRC7480_G614 at Month 2-Peru | 13 | 2 | 17 | 11 | 20 | 17 | 14
  VRC7480_G614 at Month 2-Total: number analyzed (Participants) | 27 | 8 | 38 | 33 | 34 | 30 | 46
  VRC7480_G614 at Month 2-Total | 22 | 6 | 33 | 29 | 30 | 30 | 41
  VRC7480_G614 at Month 2-USA: number analyzed (Participants) | 10 | 6 | 18 | 19 | 12 | 13 | 32
  VRC7480_G614 at Month 2-USA | 9 | 4 | 16 | 18 | 10 | 13 | 27
  VRC7480_G614 at Month 4-Peru: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 7
  VRC7480_G614 at Month 4-Peru | 1 |  | 1 |  |  |  | 7
  VRC7480_G614 at Month 4-Total: number analyzed (Participants) | 1 | 1 | 2 | 0 | 3 | 2 | 15
  VRC7480_G614 at Month 4-Total | 1 | 1 | 2 |  | 2 | 2 | 14
  VRC7480_G614 at Month 4-USA: number analyzed (Participants) | 0 | 1 | 1 | 0 | 3 | 2 | 8
  VRC7480_G614 at Month 4-USA |  | 1 | 1 |  | 2 | 2 | 7

8. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Enrollment Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2,3,4, overall and by region and enrollment group among America Cohort (USA and Peru only)
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Titer
  VRC7480_G614-ID50 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 49
  VRC7480_G614-ID50 at Month 0-Peru | 179.3 [68.2 to 399.8] | 684.8 [83.9 to 1352.6] | 328.7 [142.5 to 1377.7] | 1140.6 [712.2 to 2224.6] | 3636.2 [962.4 to 8836.3] | 2907.6 [1731 to 9196] | 910.9 [350.2 to 3607.9]
  VRC7480_G614-ID50 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 51 | 48 | 50 | 98
  VRC7480_G614-ID50 at Month 0-Total | 81.8 [10 to 267.5] | 83.2 [5 to 401.3] | 315.9 [101.6 to 1078.9] | 743.7 [225.1 to 1974.4] | 984.6 [252.4 to 4078.2] | 1801.9 [664 to 5198.6] | 518.2 [84.6 to 1916.2]
  VRC7480_G614-ID50 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 25 | 49
  VRC7480_G614-ID50 at Month 0-USA | 40.1 [5 to 105.9] | 62.2 [5 to 210] | 235.6 [101.5 to 1002.7] | 392.2 [186.6 to 1569.3] | 316.8 [100.8 to 1147.9] | 1232.5 [350.7 to 2627.8] | 130.2 [45.7 to 588.9]
  VRC7480_G614-ID50 at Month 12-Peru: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 6
  VRC7480_G614-ID50 at Month 12-Peru |  |  | 866.7 [866.7 to 866.7] |  |  |  | 204.9 [78.9 to 440.7]
  VRC7480_G614-ID50 at Month 12-Total: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 3 | 15
  VRC7480_G614-ID50 at Month 12-Total |  | 346.4 [346.4 to 346.4] | 737.7 [673.2 to 802.2] | 1034.5 [1034.5 to 1034.5] | 117.8 [117.8 to 117.8] | 430.5 [271.8 to 578.4] | 232.2 [62.7 to 350.8]
  VRC7480_G614-ID50 at Month 12-USA: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 3 | 9
  VRC7480_G614-ID50 at Month 12-USA |  | 346.4 [346.4 to 346.4] | 608.8 [608.8 to 608.8] | 1034.5 [1034.5 to 1034.5] | 117.8 [117.8 to 117.8] | 430.5 [271.8 to 578.4] | 232.2 [60.3 to 281.8]
  VRC7480_G614-ID50 at Month 2-Peru: number analyzed (Participants) | 17 | 2 | 20 | 14 | 22 | 17 | 14
  VRC7480_G614-ID50 at Month 2-Peru | 30.6 [10 to 48.3] | 167.6 [106.9 to 228.4] | 56.8 [10 to 99.6] | 154.5 [54.4 to 428.2] | 336.5 [202.3 to 650.4] | 951.8 [335.2 to 1387.5] | 301.5 [193.6 to 653.2]
  VRC7480_G614-ID50 at Month 2-Total: number analyzed (Participants) | 27 | 8 | 38 | 33 | 34 | 30 | 46
  VRC7480_G614-ID50 at Month 2-Total | 35.1 [10 to 56.2] | 48.6 [35.9 to 186.1] | 70.8 [10 to 137.9] | 204 [63.5 to 555.9] | 268.3 [65 to 703.7] | 458.1 [289.2 to 1173.5] | 139.8 [40.7 to 340.5]
  VRC7480_G614-ID50 at Month 2-USA: number analyzed (Participants) | 10 | 6 | 18 | 19 | 12 | 13 | 32
  VRC7480_G614-ID50 at Month 2-USA | 38.3 [26.1 to 78.2] | 48.6 [15.6 to 126.4] | 89.9 [44.9 to 149.6] | 282.8 [112.4 to 653.9] | 148.3 [23.9 to 802.2] | 358 [176.8 to 479.9] | 61.2 [24.4 to 225.1]
  VRC7480_G614-ID50 at Month 4-Peru: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 7
  VRC7480_G614-ID50 at Month 4-Peru | 113.2 [113.2 to 113.2] |  | 29.4 [29.4 to 29.4] |  |  |  | 232.2 [118.2 to 328.8]
  VRC7480_G614-ID50 at Month 4-Total: number analyzed (Participants) | 1 | 1 | 2 | 0 | 3 | 2 | 15
  VRC7480_G614-ID50 at Month 4-Total | 113.2 [113.2 to 113.2] | 253.3 [253.3 to 253.3] | 239.8 [134.6 to 345] |  | 120.2 [62.6 to 419.6] | 690.4 [518.4 to 862.5] | 187.1 [89.5 to 346.9]
  VRC7480_G614-ID50 at Month 4-USA: number analyzed (Participants) | 0 | 1 | 1 | 0 | 3 | 2 | 8
  VRC7480_G614-ID50 at Month 4-USA |  | 253.3 [253.3 to 253.3] | 450.2 [450.2 to 450.2] |  | 120.2 [62.6 to 419.6] | 690.4 [518.4 to 862.5] | 152.4 [85.5 to 323.3]
  VRC7480_G614-ID80 at Month 0-Peru: number analyzed (Participants) | 25 | 4 | 25 | 25 | 24 | 25 | 49
  VRC7480_G614-ID80 at Month 0-Peru | 42.5 [25.5 to 120.2] | 103.3 [26.4 to 187.3] | 80.4 [39.2 to 225.3] | 209 [105.6 to 565.1] | 587.9 [226.1 to 962] | 622.4 [531.4 to 1101.3] | 215.5 [99.1 to 842.9]
  VRC7480_G614-ID80 at Month 0-Total: number analyzed (Participants) | 49 | 22 | 53 | 51 | 48 | 50 | 98
  VRC7480_G614-ID80 at Month 0-Total | 29.1 [10 to 68.8] | 26.8 [5 to 110.9] | 56.7 [29.1 to 179.8] | 144.4 [53.5 to 517.4] | 225.8 [77.9 to 648.9] | 554.4 [172.3 to 948.7] | 130.2 [27.8 to 454.4]
  VRC7480_G614-ID80 at Month 0-USA: number analyzed (Participants) | 24 | 18 | 28 | 26 | 24 | 25 | 49
  VRC7480_G614-ID80 at Month 0-USA | 10 [5 to 34.7] | 22.1 [5 to 50.1] | 44.1 [27.9 to 145.7] | 110 [43.8 to 310] | 121.4 [31.9 to 217.4] | 240.9 [105.7 to 615.5] | 36.6 [10 to 148.5]
  VRC7480_G614-ID80 at Month 12-Peru: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 6
  VRC7480_G614-ID80 at Month 12-Peru |  |  | 259.2 [259.2 to 259.2] |  |  |  | 75.5 [46.2 to 127.6]
  VRC7480_G614-ID80 at Month 12-Total: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 3 | 15
  VRC7480_G614-ID80 at Month 12-Total |  | 120.4 [120.4 to 120.4] | 220.7 [201.4 to 239.9] | 334 [334 to 334] | 44.1 [44.1 to 44.1] | 128.3 [82.8 to 157] | 73.5 [27.5 to 123.4]
  VRC7480_G614-ID80 at Month 12-USA: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 3 | 9
  VRC7480_G614-ID80 at Month 12-USA |  | 120.4 [120.4 to 120.4] | 182.2 [182.2 to 182.2] | 334 [334 to 334] | 44.1 [44.1 to 44.1] | 128.3 [82.8 to 157] | 73.5 [24.4 to 111.5]
  VRC7480_G614-ID80 at Month 2-Peru: number analyzed (Participants) | 17 | 2 | 20 | 14 | 22 | 17 | 14
  VRC7480_G614-ID80 at Month 2-Peru | 10 [10 to 20.3] | 84.6 [53.6 to 115.5] | 25.5 [10 to 35.3] | 39.6 [23.5 to 130.4] | 129.9 [56.6 to 187.6] | 302.5 [116 to 518.7] | 124.2 [58.5 to 175.9]
  VRC7480_G614-ID80 at Month 2-Total: number analyzed (Participants) | 27 | 8 | 38 | 33 | 34 | 30 | 46
  VRC7480_G614-ID80 at Month 2-Total | 10 [10 to 23.9] | 22.6 [16.6 to 69.8] | 25.7 [10 to 36.9] | 48.7 [28.5 to 171.2] | 107.5 [26.4 to 188.1] | 159.3 [62.4 to 338.3] | 47.6 [10 to 126]
  VRC7480_G614-ID80 at Month 2-USA: number analyzed (Participants) | 10 | 6 | 18 | 19 | 12 | 13 | 32
  VRC7480_G614-ID80 at Month 2-USA | 10 [10 to 27.4] | 21.4 [8.9 to 43.3] | 26.5 [10 to 43.1] | 51 [35.4 to 182.7] | 50.6 [10 to 191.8] | 82.1 [44.8 to 172.8] | 22.9 [10 to 69.4]
  VRC7480_G614-ID80 at Month 4-Peru: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 7
  VRC7480_G614-ID80 at Month 4-Peru | 37.3 [37.3 to 37.3] |  | 13.7 [13.7 to 13.7] |  |  |  | 73.5 [43.2 to 122.9]
  VRC7480_G614-ID80 at Month 4-Total: number analyzed (Participants) | 1 | 1 | 2 | 0 | 3 | 2 | 15
  VRC7480_G614-ID80 at Month 4-Total | 37.3 [37.3 to 37.3] | 80.7 [80.7 to 80.7] | 76 [44.8 to 107.1] |  | 46.6 [25.8 to 111.8] | 227.2 [173.8 to 280.6] | 62.6 [30.6 to 119.6]
  VRC7480_G614-ID80 at Month 4-USA: number analyzed (Participants) | 0 | 1 | 1 | 0 | 3 | 2 | 8
  VRC7480_G614-ID80 at Month 4-USA |  | 80.7 [80.7 to 80.7] | 138.2 [138.2 to 138.2] |  | 46.6 [25.8 to 111.8] | 227.2 [173.8 to 280.6] | 53.4 [29.1 to 115.6]

9. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Enrollment Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and enrollment group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: The 'Overall Number of Participants Analyzed' summarized the participants number in South Africa population, regardless the assay availability. The 'Number Analyzed' for each antigen summarized the participants number at each time point with available assay data. The 'Number Analyzed' may be smaller than 'Overall Number of Participants Analyzed' due to assay data unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 79 | 17 | 129 | 26 | 73 | 24 | 24
Participants
  SARS-Cov-2 D614G at Month 0-RSA: number analyzed (Participants) | 54 | 11 | 94 | 17 | 41 | 13 | 9
  SARS-Cov-2 D614G at Month 0-RSA | 48 | 11 | 87 | 17 | 37 | 13 | 9
  SARS-Cov-2 D614G at Month 0-Total: number analyzed (Participants) | 69 | 14 | 125 | 22 | 57 | 18 | 18
  SARS-Cov-2 D614G at Month 0-Total | 59 | 14 | 110 | 22 | 51 | 18 | 18
  SARS-Cov-2 D614G at Month 0-non-RSA: number analyzed (Participants) | 15 | 3 | 31 | 5 | 16 | 5 | 9
  SARS-Cov-2 D614G at Month 0-non-RSA | 11 | 3 | 23 | 5 | 14 | 5 | 9
  SARS-Cov-2 D614G at Month 12-RSA: number analyzed (Participants) | 32 | 2 | 42 | 4 | 23 | 6 | 3
  SARS-Cov-2 D614G at Month 12-RSA | 31 | 2 | 41 | 4 | 23 | 6 | 3
  SARS-Cov-2 D614G at Month 12-Total: number analyzed (Participants) | 46 | 5 | 70 | 7 | 33 | 9 | 11
  SARS-Cov-2 D614G at Month 12-Total | 44 | 5 | 68 | 7 | 33 | 9 | 10
  SARS-Cov-2 D614G at Month 12-non-RSA: number analyzed (Participants) | 14 | 3 | 28 | 3 | 10 | 3 | 8
  SARS-Cov-2 D614G at Month 12-non-RSA | 13 | 3 | 27 | 3 | 10 | 3 | 7
  SARS-Cov-2 D614G at Month 2-RSA: number analyzed (Participants) | 36 | 4 | 65 | 10 | 28 | 8 | 7
  SARS-Cov-2 D614G at Month 2-RSA | 32 | 4 | 60 | 10 | 27 | 8 | 7
  SARS-Cov-2 D614G at Month 2-Total: number analyzed (Participants) | 51 | 7 | 95 | 13 | 44 | 12 | 15
  SARS-Cov-2 D614G at Month 2-Total | 43 | 7 | 80 | 13 | 43 | 12 | 14
  SARS-Cov-2 D614G at Month 2-non-RSA: number analyzed (Participants) | 15 | 3 | 30 | 3 | 16 | 4 | 8
  SARS-Cov-2 D614G at Month 2-non-RSA | 11 | 3 | 20 | 3 | 16 | 4 | 7
  SARS-Cov-2 D614G at Month 4-RSA: number analyzed (Participants) | 38 | 3 | 64 | 11 | 29 | 6 | 6
  SARS-Cov-2 D614G at Month 4-RSA | 34 | 3 | 58 | 10 | 27 | 6 | 6
  SARS-Cov-2 D614G at Month 4-Total: number analyzed (Participants) | 51 | 6 | 89 | 14 | 43 | 11 | 14
  SARS-Cov-2 D614G at Month 4-Total | 46 | 6 | 79 | 13 | 40 | 11 | 13
  SARS-Cov-2 D614G at Month 4-non-RSA: number analyzed (Participants) | 13 | 3 | 25 | 3 | 14 | 5 | 8
  SARS-Cov-2 D614G at Month 4-non-RSA | 12 | 3 | 21 | 3 | 13 | 5 | 7

10. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Enrollment Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and enrollment group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 79 | 17 | 129 | 26 | 73 | 24 | 24
Titer
  SARS-Cov-2 D614G-ID50 at Month 0-RSA: number analyzed (Participants) | 54 | 11 | 94 | 17 | 41 | 13 | 9
  SARS-Cov-2 D614G-ID50 at Month 0-RSA | 169 [45.7 to 350.5] | 358.7 [212.6 to 1295.5] | 303.2 [126.7 to 1449.2] | 478.7 [190.5 to 1039.8] | 501.5 [172.5 to 1157.5] | 1570.3 [947.6 to 2243.8] | 1950.5 [320.3 to 2365.9]
  SARS-Cov-2 D614G-ID50 at Month 0-Total: number analyzed (Participants) | 69 | 14 | 125 | 22 | 57 | 18 | 18
  SARS-Cov-2 D614G-ID50 at Month 0-Total | 169.6 [34.2 to 309.4] | 239.3 [153 to 723.5] | 288.3 [77.5 to 1183.3] | 761.8 [226.6 to 1071.6] | 543.4 [135 to 1560.6] | 1645.9 [994.1 to 2637.6] | 1141.3 [331.1 to 2336.7]
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA: number analyzed (Participants) | 15 | 3 | 31 | 5 | 16 | 5 | 9
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA | 183.5 [6.6 to 232.5] | 59.5 [33.9 to 74.2] | 155.4 [7.5 to 418.9] | 1149 [909.9 to 1860.1] | 971 [129.4 to 1685.7] | 2610.3 [1535.3 to 3762] | 637.8 [363.3 to 2012.3]
  SARS-Cov-2 D614G-ID50 at Month 12-RSA: number analyzed (Participants) | 32 | 2 | 42 | 4 | 23 | 6 | 3
  SARS-Cov-2 D614G-ID50 at Month 12-RSA | 312.6 [99.3 to 2118.2] | 7946.9 [7215.5 to 8678.4] | 2071.9 [405.6 to 9058.9] | 18743.3 [4428.6 to 86976.3] | 2700 [1307.3 to 11734.9] | 13387 [5435.6 to 23224.6] | 296.8 [248.8 to 2950.3]
  SARS-Cov-2 D614G-ID50 at Month 12-Total: number analyzed (Participants) | 46 | 5 | 70 | 7 | 33 | 9 | 11
  SARS-Cov-2 D614G-ID50 at Month 12-Total | 451.6 [175 to 2191.2] | 6268.4 [612.4 to 6484] | 796.8 [286.6 to 7428.8] | 5616.2 [814.7 to 19901.6] | 2443.4 [654.1 to 7211.4] | 11384.1 [3452.8 to 25836.3] | 600.5 [277.5 to 13651.4]
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA: number analyzed (Participants) | 14 | 3 | 28 | 3 | 10 | 3 | 8
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA | 1305.9 [342.3 to 2191.2] | 612.4 [362 to 3440.4] | 426.7 [225 to 1844.7] | 763.5 [595 to 4348.2] | 1657.7 [382.1 to 5252.7] | 3743.2 [1976.1 to 28947.3] | 4857.5 [283.5 to 21796.8]
  SARS-Cov-2 D614G-ID50 at Month 2-RSA: number analyzed (Participants) | 36 | 4 | 65 | 10 | 28 | 8 | 7
  SARS-Cov-2 D614G-ID50 at Month 2-RSA | 82.3 [10 to 208] | 156.4 [76.1 to 276.7] | 121 [57.8 to 518.5] | 377.4 [193 to 805.4] | 270.7 [76.7 to 823.3] | 783.2 [432.4 to 1058.8] | 627.8 [317.6 to 1373.4]
  SARS-Cov-2 D614G-ID50 at Month 2-Total: number analyzed (Participants) | 51 | 7 | 95 | 13 | 44 | 12 | 15
  SARS-Cov-2 D614G-ID50 at Month 2-Total | 68.3 [10 to 197.6] | 71.4 [53.5 to 156.4] | 95.3 [30.9 to 320.4] | 356.5 [238.6 to 726.4] | 244.6 [64.1 to 621.5] | 852.9 [477.7 to 1354] | 422 [122.5 to 1104.7]
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA: number analyzed (Participants) | 15 | 3 | 30 | 3 | 16 | 4 | 8
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA | 50.9 [7.5 to 179.6] | 52.8 [30.5 to 62.1] | 43.2 [5 to 141.6] | 356.5 [297.5 to 410.8] | 218.7 [49.4 to 404.2] | 1698.5 [769.6 to 4066.8] | 122.5 [43.3 to 946.5]
  SARS-Cov-2 D614G-ID50 at Month 4-RSA: number analyzed (Participants) | 38 | 3 | 64 | 11 | 29 | 6 | 6
  SARS-Cov-2 D614G-ID50 at Month 4-RSA | 211.1 [47.2 to 636.3] | 142.7 [109.5 to 191.7] | 323.3 [79.8 to 971.3] | 396.2 [208.6 to 900.2] | 446.4 [105.3 to 1347.6] | 772.5 [356.5 to 1276.4] | 720.4 [492.5 to 1095]
  SARS-Cov-2 D614G-ID50 at Month 4-Total: number analyzed (Participants) | 51 | 6 | 89 | 14 | 43 | 11 | 14
  SARS-Cov-2 D614G-ID50 at Month 4-Total | 163 [51.4 to 383.1] | 130.7 [86.9 to 147.1] | 252.1 [62.2 to 869.3] | 458.3 [261 to 569.4] | 450.3 [97.2 to 1132] | 954.2 [519.4 to 2129.6] | 633.8 [267.7 to 1152.3]
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA: number analyzed (Participants) | 13 | 3 | 25 | 3 | 14 | 5 | 8
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA | 135.2 [76.8 to 185.4] | 118.7 [63.5 to 133.6] | 99.2 [10 to 276.5] | 520.5 [416.5 to 538.9] | 538 [77.4 to 1126.2] | 2671.3 [954.2 to 4229] | 537.5 [172.5 to 1314]
  SARS-Cov-2 D614G-ID80 at Month 0-RSA: number analyzed (Participants) | 54 | 11 | 94 | 17 | 41 | 13 | 9
  SARS-Cov-2 D614G-ID80 at Month 0-RSA | 40.2 [10 to 117.1] | 82.2 [52.2 to 229] | 78.3 [34.4 to 340.5] | 181.5 [51.7 to 207.5] | 131.6 [37.3 to 394.4] | 572.9 [258.7 to 605.8] | 399.5 [117 to 680.3]
  SARS-Cov-2 D614G-ID80 at Month 0-Total: number analyzed (Participants) | 69 | 14 | 125 | 22 | 57 | 18 | 18
  SARS-Cov-2 D614G-ID80 at Month 0-Total | 38.7 [10 to 95.8] | 58.2 [34.5 to 212.8] | 62.8 [27.5 to 214.1] | 190.8 [59.5 to 309.7] | 138.1 [36.7 to 394.4] | 573.5 [275.7 to 609.3] | 283.5 [101.8 to 664]
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA: number analyzed (Participants) | 15 | 3 | 31 | 5 | 16 | 5 | 9
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA | 36.7 [6.3 to 49.6] | 24.7 [16.1 to 27.1] | 31.9 [7.5 to 117.6] | 274.7 [182.1 to 612.6] | 237.2 [35.3 to 438.9] | 610.4 [326.9 to 1009.9] | 167.5 [101.4 to 615.2]
  SARS-Cov-2 D614G-ID80 at Month 12-RSA: number analyzed (Participants) | 32 | 2 | 42 | 4 | 23 | 6 | 3
  SARS-Cov-2 D614G-ID80 at Month 12-RSA | 103.4 [35.4 to 719.6] | 2108.9 [1594 to 2623.7] | 605.6 [114.7 to 2737.1] | 4870.3 [990.6 to 26125.8] | 698.9 [270 to 3349.1] | 3519.1 [1372.1 to 5869] | 62.8 [59 to 720.9]
  SARS-Cov-2 D614G-ID80 at Month 12-Total: number analyzed (Participants) | 46 | 5 | 70 | 7 | 33 | 9 | 11
  SARS-Cov-2 D614G-ID80 at Month 12-Total | 135.6 [39 to 708.1] | 945.6 [161.2 to 1079.1] | 217.2 [103.5 to 1729.5] | 1237.1 [212 to 5302] | 694.1 [224 to 2500] | 3310.6 [725.9 to 6582.8] | 190.8 [81.4 to 3046.5]
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA: number analyzed (Participants) | 14 | 3 | 28 | 3 | 10 | 3 | 8
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA | 431.1 [100.5 to 673.1] | 161.2 [96.5 to 553.4] | 137.4 [65.5 to 600.9] | 173.2 [144.4 to 1136.9] | 437.3 [161.7 to 1717] | 971.6 [517.2 to 8470] | 1389.2 [117 to 5979.9]
  SARS-Cov-2 D614G-ID80 at Month 2-RSA: number analyzed (Participants) | 36 | 4 | 65 | 10 | 28 | 8 | 7
  SARS-Cov-2 D614G-ID80 at Month 2-RSA | 31.7 [10 to 47.1] | 35.1 [24.9 to 52.1] | 36.4 [10 to 139.5] | 125.7 [44.2 to 191.7] | 92.5 [31 to 228.2] | 184.8 [155.4 to 199.6] | 173.5 [87.3 to 408.7]
  SARS-Cov-2 D614G-ID80 at Month 2-Total: number analyzed (Participants) | 51 | 7 | 95 | 13 | 44 | 12 | 15
  SARS-Cov-2 D614G-ID80 at Month 2-Total | 20.9 [10 to 41.2] | 23.6 [16.2 to 35.1] | 34 [10 to 91.8] | 122.2 [43.6 to 182.3] | 89.2 [26.6 to 167.3] | 188.6 [155.4 to 224] | 105 [31.3 to 302.2]
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA: number analyzed (Participants) | 15 | 3 | 30 | 3 | 16 | 4 | 8
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA | 10 [6.3 to 29.6] | 22.5 [15 to 23.1] | 10 [5 to 37.8] | 122.2 [82.9 to 136.6] | 74.1 [12.2 to 119.7] | 351.7 [162.8 to 797] | 31.3 [21.4 to 259.4]
  SARS-Cov-2 D614G-ID80 at Month 4-RSA: number analyzed (Participants) | 38 | 3 | 64 | 11 | 29 | 6 | 6
  SARS-Cov-2 D614G-ID80 at Month 4-RSA | 51.9 [10 to 163.8] | 31.9 [27.3 to 32.9] | 100.9 [26.1 to 236.5] | 101 [40.4 to 214.2] | 121.9 [37.6 to 408.7] | 190.4 [92.3 to 441.3] | 164.2 [141.4 to 251.4]
  SARS-Cov-2 D614G-ID80 at Month 4-Total: number analyzed (Participants) | 51 | 6 | 89 | 14 | 43 | 11 | 14
  SARS-Cov-2 D614G-ID80 at Month 4-Total | 42.1 [10 to 130.8] | 32.9 [25 to 33.8] | 66.6 [21.8 to 206.1] | 116.4 [55.4 to 182.5] | 124 [33.7 to 288.9] | 234.7 [151.2 to 674.6] | 164.2 [65.9 to 286.1]
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA: number analyzed (Participants) | 13 | 3 | 25 | 3 | 14 | 5 | 8
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA | 34.2 [26.6 to 43.3] | 33.8 [20.7 to 36.3] | 36.4 [10 to 89.2] | 147.3 [133.3 to 168.1] | 163.9 [29.8 to 276.1] | 717.7 [234.7 to 749.6] | 144.5 [45.6 to 386.7]

11. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (ADCC) by Region and Enrollment Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by antibody-dependent cellular cytotoxicity assay (ADCC) at Visit 1, overall and by region and enrollment group among America Cohort (USA and Peru only)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 7: Clinical spectrums , age 18 - 55
- Group 8: Clinical spectrums , age 55+
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 81 | 20
Participants
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru: number analyzed (Participants) | 20 | 4 | 19 | 17 | 21 | 17 | 24 | 6
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru | 8 | 2 | 11 | 13 | 17 | 17 | 19 | 5
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 36 | 20 | 30 | 33 | 35 | 35 | 49 | 18
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 10 | 4 | 14 | 22 | 28 | 33 | 29 | 12
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA: number analyzed (Participants) | 16 | 16 | 11 | 16 | 14 | 18 | 25 | 12
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA | 2 | 2 | 3 | 9 | 11 | 16 | 10 | 7
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru: number analyzed (Participants) | 20 | 4 | 19 | 17 | 21 | 17 | 24 | 6
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru | 7 | 3 | 13 | 13 | 18 | 16 | 19 | 6
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 36 | 20 | 30 | 33 | 35 | 35 | 49 | 18
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 9 | 6 | 20 | 21 | 27 | 27 | 30 | 13
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA: number analyzed (Participants) | 16 | 16 | 11 | 16 | 14 | 18 | 25 | 12
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA | 2 | 3 | 7 | 8 | 9 | 11 | 11 | 7

12. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (ADCC) by Region and Enrollment Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by antibody-dependent cellular cytotoxicity assay (ADCC) Visit 1, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: Percent CD107a+ NK Cells
Groups:
- Group 2: Asymptomatic, age > 55
- Group 4: Symptomatic, age > 55
- Group 6: Hospitalized, age > 55
- Group 8: Clinical spectrums , age > 55
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 81 | 20
Percent CD107a+ NK Cells
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru: number analyzed (Participants) | 20 | 4 | 19 | 17 | 21 | 17 | 24 | 6
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru | 1.5 [0.5 to 4.4] | 3.7 [1.1 to 6.3] | 5 [1.9 to 13.8] | 8.8 [4.5 to 15.1] | 12.6 [6.5 to 14.9] | 13.6 [12.4 to 20.9] | 8.9 [5.3 to 17.3] | 15.5 [11.6 to 22.4]
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 36 | 20 | 30 | 33 | 35 | 35 | 49 | 18
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 1.2 [0 to 4.1] | 0.8 [0 to 2.6] | 3.4 [1 to 9.4] | 6.5 [3.5 to 11.8] | 10.8 [4.6 to 14.8] | 14.1 [11.6 to 18.8] | 6.3 [2.1 to 14] | 10.8 [2 to 16]
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA: number analyzed (Participants) | 16 | 16 | 11 | 16 | 14 | 18 | 25 | 12
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA | 1 [0 to 2.1] | 0.3 [0 to 2] | 1.4 [0.3 to 3.9] | 4.6 [3.5 to 7.8] | 7.7 [4.3 to 13.3] | 15.3 [10 to 18.1] | 3.3 [1.1 to 7.5] | 6.7 [1.6 to 12.9]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru: number analyzed (Participants) | 20 | 4 | 19 | 17 | 21 | 17 | 24 | 6
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru | 4.5 [2.2 to 8] | 8.3 [4.3 to 11.8] | 8 [3.6 to 12.3] | 8.6 [5.3 to 11.3] | 15.7 [11.4 to 18] | 15.2 [12.6 to 18.7] | 9.8 [6.6 to 14.3] | 16.5 [15.1 to 16.8]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 36 | 20 | 30 | 33 | 35 | 35 | 49 | 18
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 3.4 [0.5 to 5.3] | 2.8 [0 to 5.9] | 6.7 [4.1 to 12.4] | 6.8 [3.8 to 10.2] | 13.1 [7.2 to 16.9] | 12.5 [5.8 to 15.6] | 6.8 [3.6 to 11.2] | 8.8 [4.7 to 15.2]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA: number analyzed (Participants) | 16 | 16 | 11 | 16 | 14 | 18 | 25 | 12
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA | 1.4 [0 to 4.3] | 1.4 [0 to 4.7] | 5.6 [4.2 to 9.9] | 5.8 [2.7 to 8.8] | 9.4 [3.3 to 13] | 7.7 [2.8 to 12.3] | 4.5 [2.8 to 8.2] | 5.8 [3.5 to 8.6]

13. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate (ICS) by Region and Enrollment Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate by flow cytometry at Visit 1 , overall and by region and enrollment group among America Cohort (USA and Peru only)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 1B: 1B: Asymptomatic, 55+
- Group 1D: 1D: Symptomatic, 55+
- Group 2B: 2B: Hospitalized, 55+
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD4+-Any COV2 at Month 0-Peru | 12 | 3 | 13 | 23 | 20 | 25 | 47
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 48 | 21 | 53 | 50 | 48 | 49 | 96
  CD4+-Any COV2 at Month 0-Total | 21 | 11 | 31 | 46 | 37 | 47 | 79
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 28 | 25 | 24 | 24 | 47
  CD4+-Any COV2 at Month 0-USA | 9 | 8 | 18 | 23 | 17 | 22 | 32
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 25 | 25 | 24 | 25 | 48
  CD4+-E M at Month 0-Peru | 5 | 2 | 9 | 20 | 17 | 22 | 40
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 46 | 20 | 53 | 49 | 48 | 48 | 94
  CD4+-E M at Month 0-Total | 10 | 5 | 20 | 40 | 32 | 39 | 57
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 23 | 16 | 28 | 24 | 24 | 23 | 46
  CD4+-E M at Month 0-USA | 5 | 3 | 11 | 20 | 15 | 17 | 17
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD4+-N at Month 0-Peru | 9 | 2 | 10 | 21 | 16 | 21 | 37
  CD4+-N at Month 0-Total: number analyzed (Participants) | 48 | 20 | 53 | 50 | 48 | 49 | 96
  CD4+-N at Month 0-Total | 14 | 5 | 24 | 44 | 30 | 43 | 61
  CD4+-N at Month 0-USA: number analyzed (Participants) | 24 | 16 | 28 | 25 | 24 | 24 | 47
  CD4+-N at Month 0-USA | 5 | 3 | 14 | 23 | 14 | 22 | 24
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 24 | 24 | 25 | 46
  CD4+-ORF3a6 at Month 0-Peru | 1 | 2 | 3 | 17 | 9 | 12 | 21
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 47 | 20 | 53 | 49 | 48 | 48 | 92
  CD4+-ORF3a6 at Month 0-Total | 3 | 5 | 7 | 29 | 22 | 29 | 31
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 23 | 16 | 28 | 25 | 24 | 23 | 46
  CD4+-ORF3a6 at Month 0-USA | 2 | 3 | 4 | 12 | 13 | 17 | 10
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 47
  CD4+-ORF7a7b8 at Month 0-Peru | 3 | 2 | 4 | 17 | 12 | 19 | 29
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 47 | 19 | 52 | 49 | 48 | 47 | 94
  CD4+-ORF7a7b8 at Month 0-Total | 3 | 5 | 8 | 30 | 21 | 32 | 43
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 23 | 15 | 27 | 24 | 24 | 22 | 47
  CD4+-ORF7a7b8 at Month 0-USA | 0 | 3 | 4 | 13 | 9 | 13 | 14
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 25 | 25 | 24 | 24 | 48
  CD4+-S1 at Month 0-Peru | 8 | 2 | 12 | 20 | 19 | 24 | 41
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 47 | 21 | 53 | 50 | 47 | 48 | 95
  CD4+-S1 at Month 0-Total | 12 | 7 | 25 | 41 | 35 | 45 | 66
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 28 | 25 | 23 | 24 | 47
  CD4+-S1 at Month 0-USA | 4 | 5 | 13 | 21 | 16 | 21 | 25
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD4+-S2 at Month 0-Peru | 10 | 2 | 7 | 18 | 16 | 24 | 39
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 48 | 21 | 53 | 50 | 48 | 49 | 96
  CD4+-S2 at Month 0-Total | 13 | 8 | 19 | 37 | 32 | 45 | 65
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 28 | 25 | 24 | 24 | 47
  CD4+-S2 at Month 0-USA | 3 | 6 | 12 | 19 | 16 | 21 | 26
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD4+-Spike at Month 0-Peru | 11 | 2 | 12 | 20 | 20 | 25 | 45
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 48 | 21 | 53 | 50 | 48 | 49 | 96
  CD4+-Spike at Month 0-Total | 16 | 8 | 27 | 43 | 37 | 46 | 75
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 24 | 17 | 28 | 25 | 24 | 24 | 47
  CD4+-Spike at Month 0-USA | 5 | 6 | 15 | 23 | 17 | 21 | 30
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD8+-Any COV2 at Month 0-Peru | 13 | 1 | 17 | 18 | 19 | 19 | 35
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 48 | 21 | 52 | 50 | 48 | 49 | 96
  CD8+-Any COV2 at Month 0-Total | 23 | 8 | 33 | 37 | 35 | 33 | 63
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 27 | 25 | 24 | 24 | 47
  CD8+-Any COV2 at Month 0-USA | 10 | 7 | 16 | 19 | 16 | 14 | 28
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 48
  CD8+-E M at Month 0-Peru | 0 | 0 | 0 | 1 | 2 | 3 | 7
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 47 | 20 | 52 | 49 | 48 | 48 | 94
  CD8+-E M at Month 0-Total | 1 | 1 | 3 | 5 | 3 | 7 | 10
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 23 | 16 | 27 | 24 | 24 | 23 | 46
  CD8+-E M at Month 0-USA | 1 | 1 | 3 | 4 | 1 | 4 | 3
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD8+-N at Month 0-Peru | 10 | 1 | 15 | 18 | 17 | 16 | 31
  CD8+-N at Month 0-Total: number analyzed (Participants) | 48 | 20 | 52 | 50 | 48 | 49 | 96
  CD8+-N at Month 0-Total | 19 | 7 | 26 | 36 | 31 | 26 | 55
  CD8+-N at Month 0-USA: number analyzed (Participants) | 24 | 16 | 27 | 25 | 24 | 24 | 47
  CD8+-N at Month 0-USA | 9 | 6 | 11 | 18 | 14 | 10 | 24
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 47
  CD8+-ORF3a6 at Month 0-Peru | 4 | 0 | 6 | 8 | 11 | 7 | 14
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 47 | 20 | 52 | 50 | 48 | 48 | 93
  CD8+-ORF3a6 at Month 0-Total | 6 | 2 | 8 | 14 | 15 | 13 | 22
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 23 | 16 | 27 | 25 | 24 | 23 | 46
  CD8+-ORF3a6 at Month 0-USA | 2 | 2 | 2 | 6 | 4 | 6 | 8
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 47
  CD8+-ORF7a7b8 at Month 0-Peru | 3 | 0 | 6 | 9 | 11 | 8 | 14
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 46 | 19 | 51 | 49 | 48 | 47 | 94
  CD8+-ORF7a7b8 at Month 0-Total | 5 | 0 | 6 | 14 | 15 | 11 | 20
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 22 | 15 | 26 | 24 | 24 | 22 | 47
  CD8+-ORF7a7b8 at Month 0-USA | 2 | 0 | 0 | 5 | 4 | 3 | 6
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 23 | 4 | 25 | 25 | 24 | 24 | 49
  CD8+-S1 at Month 0-Peru | 1 | 0 | 5 | 8 | 7 | 6 | 15
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 47 | 21 | 52 | 50 | 47 | 48 | 96
  CD8+-S1 at Month 0-Total | 1 | 0 | 13 | 15 | 11 | 10 | 21
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 27 | 25 | 23 | 24 | 47
  CD8+-S1 at Month 0-USA | 0 | 0 | 8 | 7 | 4 | 4 | 6
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 24 | 49
  CD8+-S2 at Month 0-Peru | 3 | 0 | 1 | 3 | 4 | 2 | 5
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 48 | 21 | 52 | 50 | 48 | 48 | 96
  CD8+-S2 at Month 0-Total | 4 | 0 | 4 | 5 | 6 | 3 | 8
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 24 | 17 | 27 | 25 | 24 | 24 | 47
  CD8+-S2 at Month 0-USA | 1 | 0 | 3 | 2 | 2 | 1 | 3
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 24 | 4 | 25 | 25 | 24 | 25 | 49
  CD8+-Spike at Month 0-Peru | 4 | 0 | 5 | 9 | 7 | 6 | 16
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 48 | 21 | 52 | 50 | 48 | 49 | 96
  CD8+-Spike at Month 0-Total | 5 | 0 | 15 | 17 | 12 | 10 | 23
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 24 | 17 | 27 | 25 | 24 | 24 | 47
  CD8+-Spike at Month 0-USA | 1 | 0 | 10 | 8 | 5 | 4 | 7

14. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude (ICS) by Region and Enrollment Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and enrollment group among America Cohort positive responders (USA and Peru)
Time Frame: Measured at Months 0
Population: American Population among positive responders (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: % T cells expressing IFN-g/IL-2
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
% T cells expressing IFN-g/IL-2
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 12 | 3 | 13 | 23 | 20 | 25 | 47
  CD4+-Any COV2 at Month 0-Peru | 0.2 [0.2 to 0.4] | 0.4 [0.2 to 0.5] | 0.4 [0.3 to 0.6] | 0.9 [0.6 to 1.4] | 0.6 [0.4 to 1.1] | 1 [0.6 to 1.5] | 0.9 [0.5 to 1.6]
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 21 | 11 | 31 | 46 | 37 | 47 | 79
  CD4+-Any COV2 at Month 0-Total | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.7] | 0.3 [0.3 to 0.6] | 0.8 [0.4 to 1.2] | 0.6 [0.4 to 1.1] | 1 [0.6 to 1.5] | 0.7 [0.3 to 1.2]
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 9 | 8 | 18 | 23 | 17 | 22 | 32
  CD4+-Any COV2 at Month 0-USA | 0.4 [0.2 to 0.4] | 0.2 [0.1 to 0.6] | 0.3 [0.2 to 0.4] | 0.6 [0.4 to 1.1] | 0.6 [0.5 to 1] | 1 [0.6 to 1.4] | 0.5 [0.3 to 0.9]
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 5 | 2 | 9 | 20 | 17 | 22 | 40
  CD4+-E M at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4]
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 10 | 5 | 20 | 40 | 32 | 39 | 57
  CD4+-E M at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 5 | 3 | 11 | 20 | 15 | 17 | 17
  CD4+-E M at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 9 | 2 | 10 | 21 | 16 | 21 | 37
  CD4+-N at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-Total: number analyzed (Participants) | 14 | 5 | 24 | 44 | 30 | 43 | 61
  CD4+-N at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-USA: number analyzed (Participants) | 5 | 3 | 14 | 23 | 14 | 22 | 24
  CD4+-N at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 1 | 2 | 3 | 17 | 9 | 12 | 21
  CD4+-ORF3a6 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 3 | 5 | 7 | 29 | 22 | 29 | 31
  CD4+-ORF3a6 at Month 0-Total | 0.4 [0.3 to 0.9] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 2 | 3 | 4 | 12 | 13 | 17 | 10
  CD4+-ORF3a6 at Month 0-USA | 0.9 [0.7 to 1.1] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.5] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 3 | 2 | 4 | 17 | 12 | 19 | 29
  CD4+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 3 | 5 | 8 | 30 | 21 | 32 | 43
  CD4+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 0 | 3 | 4 | 13 | 9 | 13 | 14
  CD4+-ORF7a7b8 at Month 0-USA |  | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 8 | 2 | 12 | 20 | 19 | 24 | 41
  CD4+-S1 at Month 0-Peru | 0.1 [0 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.5]
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 12 | 7 | 25 | 41 | 35 | 45 | 66
  CD4+-S1 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.4]
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 4 | 5 | 13 | 21 | 16 | 21 | 25
  CD4+-S1 at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.2 [0.2 to 0.4] | 0.1 [0.1 to 0.3]
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 10 | 2 | 7 | 18 | 16 | 24 | 39
  CD4+-S2 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 13 | 8 | 19 | 37 | 32 | 45 | 65
  CD4+-S2 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3]
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 3 | 6 | 12 | 19 | 16 | 21 | 26
  CD4+-S2 at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 11 | 2 | 12 | 20 | 20 | 25 | 45
  CD4+-Spike at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.3 [0.2 to 0.4] | 0.2 [0.2 to 0.3] | 0.4 [0.3 to 0.7] | 0.3 [0.1 to 0.5] | 0.4 [0.2 to 0.6] | 0.4 [0.2 to 0.8]
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 16 | 8 | 27 | 43 | 37 | 46 | 75
  CD4+-Spike at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.5] | 0.4 [0.3 to 0.6] | 0.3 [0.2 to 0.6]
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 5 | 6 | 15 | 23 | 17 | 21 | 30
  CD4+-Spike at Month 0-USA | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.7] | 0.2 [0.1 to 0.4]
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 13 | 1 | 17 | 18 | 19 | 19 | 35
  CD8+-Any COV2 at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.3 [0.3 to 0.3] | 0.5 [0.2 to 0.6] | 0.6 [0.4 to 2] | 0.9 [0.3 to 1.7] | 0.6 [0.2 to 3.8] | 0.5 [0.3 to 1.2]
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 23 | 8 | 33 | 37 | 35 | 33 | 63
  CD8+-Any COV2 at Month 0-Total | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.6] | 0.6 [0.3 to 1.5] | 0.5 [0.2 to 1.6] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 0.9]
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 10 | 7 | 16 | 19 | 16 | 14 | 28
  CD8+-Any COV2 at Month 0-USA | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.3] | 0.6 [0.3 to 1.5] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.4 [0.2 to 0.7]
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 3 | 7
  CD8+-E M at Month 0-Peru |  |  |  | 0.1 [0.1 to 0.1] | 0.2 [0.2 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 1 | 1 | 3 | 5 | 3 | 7 | 10
  CD8+-E M at Month 0-Total | 2.3 [2.3 to 2.3] | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.4] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3]
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 1 | 1 | 3 | 4 | 1 | 4 | 3
  CD8+-E M at Month 0-USA | 2.3 [2.3 to 2.3] | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.7 [0.7 to 0.7] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.4]
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 10 | 1 | 15 | 18 | 17 | 16 | 31
  CD8+-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.5] | 0.5 [0.1 to 1] | 0.4 [0.2 to 3.5] | 0.2 [0.1 to 0.6]
  CD8+-N at Month 0-Total: number analyzed (Participants) | 19 | 7 | 26 | 36 | 31 | 26 | 55
  CD8+-N at Month 0-Total | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0.3 [0.1 to 0.9] | 0.3 [0.1 to 1] | 0.2 [0.1 to 0.4]
  CD8+-N at Month 0-USA: number analyzed (Participants) | 9 | 6 | 11 | 18 | 14 | 10 | 24
  CD8+-N at Month 0-USA | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.5] | 0.1 [0.1 to 0.3]
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 4 | 0 | 6 | 8 | 11 | 7 | 14
  CD8+-ORF3a6 at Month 0-Peru | 0.1 [0.1 to 0.2] |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.9 [0.5 to 1.3] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 6 | 2 | 8 | 14 | 15 | 13 | 22
  CD8+-ORF3a6 at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.3 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.9] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 2 | 2 | 2 | 6 | 4 | 6 | 8
  CD8+-ORF3a6 at Month 0-USA | 0.3 [0.2 to 0.5] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.3 [0.3 to 0.4] | 0.3 [0.2 to 0.4] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 3 | 0 | 6 | 9 | 11 | 8 | 14
  CD8+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.2] |  | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.7] | 1 [0.5 to 2] | 0.2 [0.1 to 0.4]
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 5 | 0 | 6 | 14 | 15 | 11 | 20
  CD8+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.3] |  | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.5] | 0.3 [0.1 to 0.7] | 0.6 [0.3 to 1.6] | 0.2 [0.1 to 0.4]
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 2 | 0 | 0 | 5 | 4 | 3 | 6
  CD8+-ORF7a7b8 at Month 0-USA | 0.4 [0.2 to 0.6] |  |  | 0.1 [0.1 to 0.4] | 0.3 [0.1 to 0.6] | 0.3 [0.2 to 0.5] | 0.1 [0.1 to 0.2]
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 1 | 0 | 5 | 8 | 7 | 6 | 15
  CD8+-S1 at Month 0-Peru | 0 [0 to 0] |  | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 1 | 0 | 13 | 15 | 11 | 10 | 21
  CD8+-S1 at Month 0-Total | 0 [0 to 0] |  | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 0 | 0 | 8 | 7 | 4 | 4 | 6
  CD8+-S1 at Month 0-USA |  |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 3 | 0 | 1 | 3 | 4 | 2 | 5
  CD8+-S2 at Month 0-Peru | 0.1 [0.1 to 0.1] |  | 0.4 [0.4 to 0.4] | 0.9 [0.5 to 1.9] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2]
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 4 | 0 | 4 | 5 | 6 | 3 | 8
  CD8+-S2 at Month 0-Total | 0.1 [0.1 to 0.1] |  | 0.1 [0.1 to 0.2] | 0.6 [0.3 to 0.9] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2]
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 1 | 0 | 3 | 2 | 2 | 1 | 3
  CD8+-S2 at Month 0-USA | 0.2 [0.2 to 0.2] |  | 0.1 [0.1 to 0.1] | 0.4 [0.4 to 0.5] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.5]
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 4 | 0 | 5 | 9 | 7 | 6 | 16
  CD8+-Spike at Month 0-Peru | 0.1 [0.1 to 0.1] |  | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.5] | 0.3 [0.1 to 0.6] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 5 | 0 | 15 | 17 | 12 | 10 | 23
  CD8+-Spike at Month 0-Total | 0.1 [0.1 to 0.1] |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 1 | 0 | 10 | 8 | 5 | 4 | 7
  CD8+-Spike at Month 0-USA | 0.2 [0.2 to 0.2] |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.8] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.3 [0.2 to 0.6]

15. Primary Outcome: SARS-CoV-2-specific Memory B Cell Response Magnitude (B Cell) by Region and Enrollment Group Among America Cohort
Description: SARS-CoV-2-specific B cell responses and B cell phenotypic data was identified and characterized using fluorescently-labelled recombinant Env proteins (S6P and RBD) in combination with a flow cytometry antibody panel on all available samples from the enrollment visit (V1). There is no positivity call for B cell phenotypic data. The magnitude is B cell subset frequency.
  The table summarized SARS-CoV-2-specific Memory B Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and enrollment group among America Cohort (USA and Peru only)
Time Frame: Measured at Months 0.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
percentage of cells
  %RBD+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %RBD+ IgA+ of Memory B Cells-Peru | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.03] | 0 [0 to 0.02] | 0.04 [0.01 to 0.08] | 0.01 [0 to 0.03] | 0.03 [0.01 to 0.08] | 0 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %RBD+ IgA+ of Memory B Cells-Total | 0.01 [0 to 0.04] | 0 [0 to 0.02] | 0 [0 to 0.01] | 0.02 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.05] | 0.01 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %RBD+ IgA+ of Memory B Cells-USA | 0 [0 to 0.07] | 0 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.05] | 0 [0 to 0.02] | 0.01 [0 to 0.04]
  %RBD+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %RBD+ IgG+ of Memory B Cells-Peru | 0.08 [0.04 to 0.15] | 0.23 [0.04 to 0.41] | 0.1 [0.04 to 0.17] | 0.25 [0.1 to 0.75] | 0.14 [0.08 to 0.29] | 0.28 [0.13 to 0.45] | 0.18 [0.12 to 0.32]
  %RBD+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %RBD+ IgG+ of Memory B Cells-Total | 0.07 [0.01 to 0.15] | 0.09 [0 to 0.28] | 0.12 [0.05 to 0.2] | 0.24 [0.09 to 0.49] | 0.16 [0.08 to 0.33] | 0.28 [0.12 to 0.41] | 0.16 [0.1 to 0.3]
  %RBD+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %RBD+ IgG+ of Memory B Cells-USA | 0.06 [0 to 0.16] | 0.09 [0 to 0.26] | 0.15 [0.06 to 0.22] | 0.21 [0.08 to 0.4] | 0.21 [0.08 to 0.42] | 0.25 [0.1 to 0.37] | 0.12 [0.05 to 0.23]
  %RBD+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %RBD+ IgM+ of Memory B Cells-Peru | 0.01 [0 to 0.02] | 0 [0 to 0.02] | 0 [0 to 0] | 0.02 [0 to 0.11] | 0 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %RBD+ IgM+ of Memory B Cells-Total | 0 [0 to 0.02] | 0 [0 to 0.03] | 0 [0 to 0.01] | 0 [0 to 0.04] | 0 [0 to 0.01] | 0 [0 to 0.02] | 0 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %RBD+ IgM+ of Memory B Cells-USA | 0 [0 to 0.04] | 0 [0 to 0.03] | 0.01 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0.02] | 0 [0 to 0.02]
  %RBD+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %RBD+ of Total B Cells-Peru | 0.05 [0.04 to 0.07] | 0.05 [0.01 to 0.13] | 0.06 [0.04 to 0.08] | 0.14 [0.07 to 0.65] | 0.06 [0.04 to 0.1] | 0.11 [0.07 to 0.19] | 0.1 [0.07 to 0.14]
  %RBD+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %RBD+ of Total B Cells-Total | 0.05 [0.02 to 0.1] | 0.07 [0.03 to 0.12] | 0.05 [0.04 to 0.08] | 0.1 [0.04 to 0.14] | 0.07 [0.04 to 0.11] | 0.07 [0.05 to 0.12] | 0.07 [0.04 to 0.12]
  %RBD+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %RBD+ of Total B Cells-USA | 0.04 [0.01 to 0.21] | 0.07 [0.04 to 0.12] | 0.05 [0.04 to 0.06] | 0.07 [0.04 to 0.1] | 0.09 [0.02 to 0.17] | 0.06 [0.03 to 0.07] | 0.04 [0.03 to 0.06]
  %S+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgA+ of Memory B Cells-Peru | 0.06 [0.03 to 0.1] | 0.05 [0.02 to 0.08] | 0.08 [0.03 to 0.11] | 0.08 [0.05 to 0.12] | 0.05 [0.03 to 0.12] | 0.11 [0.05 to 0.38] | 0.07 [0.03 to 0.12]
  %S+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgA+ of Memory B Cells-Total | 0.06 [0.02 to 0.1] | 0.04 [0.01 to 0.07] | 0.06 [0.03 to 0.11] | 0.07 [0.03 to 0.12] | 0.06 [0.03 to 0.1] | 0.07 [0.02 to 0.16] | 0.08 [0.04 to 0.12]
  %S+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgA+ of Memory B Cells-USA | 0.04 [0.02 to 0.1] | 0.04 [0 to 0.05] | 0.04 [0.03 to 0.1] | 0.06 [0.02 to 0.08] | 0.07 [0.04 to 0.09] | 0.04 [0.01 to 0.08] | 0.08 [0.06 to 0.12]
  %S+ IgA+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgA+ of Total B Cells-Peru | 0.02 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.01 [0.01 to 0.02] | 0.04 [0.02 to 0.06] | 0.02 [0.01 to 0.03]
  %S+ IgA+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgA+ of Total B Cells-Total | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.03] | 0.01 [0.01 to 0.03]
  %S+ IgA+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgA+ of Total B Cells-USA | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.02 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0.01 to 0.02]
  %S+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgG+ of Memory B Cells-Peru | 0.4 [0.2 to 0.6] | 0.38 [0.27 to 0.69] | 0.43 [0.19 to 0.99] | 0.81 [0.49 to 1.12] | 0.88 [0.44 to 1.23] | 1.21 [0.85 to 1.58] | 0.83 [0.61 to 1.28]
  %S+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgG+ of Memory B Cells-Total | 0.32 [0.1 to 0.52] | 0.35 [0.04 to 0.98] | 0.49 [0.24 to 0.93] | 0.93 [0.49 to 1.55] | 0.94 [0.42 to 1.29] | 1.21 [0.71 to 1.73] | 0.7 [0.5 to 1.14]
  %S+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgG+ of Memory B Cells-USA | 0.18 [0.05 to 0.44] | 0.33 [0.04 to 0.98] | 0.69 [0.3 to 0.81] | 0.99 [0.52 to 1.69] | 1.01 [0.33 to 1.44] | 1.25 [0.62 to 1.9] | 0.58 [0.34 to 0.97]
  %S+ IgG+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgG+ of Total B Cells-Peru | 0.09 [0.05 to 0.15] | 0.04 [0.03 to 0.09] | 0.1 [0.05 to 0.21] | 0.23 [0.1 to 0.3] | 0.18 [0.1 to 0.25] | 0.26 [0.17 to 0.41] | 0.22 [0.16 to 0.29]
  %S+ IgG+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgG+ of Total B Cells-Total | 0.06 [0.02 to 0.13] | 0.05 [0.01 to 0.15] | 0.1 [0.06 to 0.19] | 0.22 [0.1 to 0.27] | 0.19 [0.09 to 0.25] | 0.19 [0.12 to 0.27] | 0.16 [0.08 to 0.24]
  %S+ IgG+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgG+ of Total B Cells-USA | 0.04 [0.01 to 0.11] | 0.11 [0 to 0.15] | 0.1 [0.07 to 0.14] | 0.18 [0.11 to 0.26] | 0.22 [0.09 to 0.26] | 0.18 [0.09 to 0.21] | 0.1 [0.05 to 0.14]
  %S+ IgM+ IgD+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgM+ IgD+ of Total B Cells-Peru | 0.12 [0.09 to 0.14] | 0.06 [0.04 to 0.09] | 0.13 [0.1 to 0.18] | 0.14 [0.11 to 0.17] | 0.11 [0.08 to 0.14] | 0.09 [0.08 to 0.14] | 0.1 [0.08 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgM+ IgD+ of Total B Cells-Total | 0.1 [0.06 to 0.13] | 0.07 [0.05 to 0.1] | 0.12 [0.09 to 0.16] | 0.13 [0.07 to 0.16] | 0.11 [0.08 to 0.15] | 0.09 [0.07 to 0.14] | 0.1 [0.07 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgM+ IgD+ of Total B Cells-USA | 0.08 [0.05 to 0.1] | 0.07 [0.05 to 0.1] | 0.1 [0.08 to 0.11] | 0.08 [0.07 to 0.13] | 0.12 [0.08 to 0.17] | 0.09 [0.05 to 0.15] | 0.09 [0.07 to 0.12]
  %S+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgM+ of Memory B Cells-Peru | 0.03 [0 to 0.08] | 0.03 [0.01 to 0.06] | 0.04 [0.02 to 0.11] | 0.06 [0.03 to 0.11] | 0.04 [0.02 to 0.06] | 0.05 [0.02 to 0.07] | 0.04 [0 to 0.06]
  %S+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgM+ of Memory B Cells-Total | 0.03 [0 to 0.09] | 0.01 [0 to 0.06] | 0.05 [0.02 to 0.08] | 0.05 [0.03 to 0.11] | 0.04 [0.01 to 0.06] | 0.05 [0.02 to 0.08] | 0.04 [0.02 to 0.08]
  %S+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgM+ of Memory B Cells-USA | 0.04 [0.01 to 0.09] | 0.01 [0 to 0.04] | 0.05 [0.03 to 0.06] | 0.04 [0.01 to 0.08] | 0.02 [0 to 0.06] | 0.04 [0.01 to 0.08] | 0.05 [0.02 to 0.08]
  %S+ IgM+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ IgM+ of Total B Cells-Peru | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.04] | 0.01 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ IgM+ of Total B Cells-Total | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.03] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ IgM+ of Total B Cells-USA | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0 [0 to 0.01] | 0 [0 to 0.01] | 0.01 [0 to 0.02]
  %S+ of Total B Cells-Peru: number analyzed (Participants) | 20 | 4 | 19 | 18 | 21 | 18 | 46
  %S+ of Total B Cells-Peru | 0.3 [0.18 to 0.37] | 0.17 [0.09 to 0.27] | 0.33 [0.24 to 0.55] | 0.51 [0.3 to 0.65] | 0.37 [0.31 to 0.52] | 0.47 [0.4 to 0.7] | 0.43 [0.32 to 0.53]
  %S+ of Total B Cells-Total: number analyzed (Participants) | 39 | 21 | 32 | 34 | 40 | 38 | 87
  %S+ of Total B Cells-Total | 0.21 [0.16 to 0.33] | 0.23 [0.1 to 0.34] | 0.28 [0.21 to 0.49] | 0.43 [0.25 to 0.57] | 0.39 [0.3 to 0.54] | 0.4 [0.28 to 0.51] | 0.35 [0.24 to 0.49]
  %S+ of Total B Cells-USA: number analyzed (Participants) | 19 | 17 | 13 | 16 | 19 | 20 | 41
  %S+ of Total B Cells-USA | 0.21 [0.11 to 0.32] | 0.24 [0.1 to 0.34] | 0.26 [0.19 to 0.34] | 0.34 [0.23 to 0.49] | 0.42 [0.3 to 0.58] | 0.3 [0.23 to 0.41] | 0.25 [0.2 to 0.35]

16. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG1) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3 , overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2, 4
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Asymptomatic
- Group 2: Symptomatic, not hospitalized
- Group 3: Hospitalized, no supp oxygen
- Group 4: Hospitalized, oxygen, no intubation/ICU
- Group 5: Hospitalized, intubation/ICU
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 15 | 41 | 27
  2019-nCoV S/293F-50 at Month 0-Peru | 18 | 46 | 15 | 41 | 27
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 53 | 106 | 19 | 62 | 44
  2019-nCoV S/293F-50 at Month 0-Total | 39 | 103 | 19 | 60 | 43
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 32 | 58 | 4 | 21 | 17
  2019-nCoV S/293F-50 at Month 0-USA | 21 | 57 | 4 | 19 | 16
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 25 | 46 | 17 | 31 | 20
  2019-nCoV S/293F-50 at Month 2-Peru | 23 | 43 | 15 | 31 | 20
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 47 | 114 | 21 | 55 | 35
  2019-nCoV S/293F-50 at Month 2-Total | 39 | 106 | 19 | 52 | 34
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 22 | 68 | 4 | 24 | 15
  2019-nCoV S/293F-50 at Month 2-USA | 16 | 63 | 4 | 21 | 14
  2019-nCoV S/293F-50 at Month 4-Peru: number analyzed (Participants) | 26 | 37 | 16 | 22 | 14
  2019-nCoV S/293F-50 at Month 4-Peru | 24 | 33 | 14 | 22 | 14
  2019-nCoV S/293F-50 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 41 | 25
  2019-nCoV S/293F-50 at Month 4-Total | 32 | 73 | 16 | 38 | 24
  2019-nCoV S/293F-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 19 | 11
  2019-nCoV S/293F-50 at Month 4-USA | 8 | 40 | 2 | 16 | 10
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 28 | 60 | 18 | 41 | 27
  SARS-CoV-2 DB His-50 at Month 0-Peru | 24 | 55 | 16 | 41 | 27
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 72 | 148 | 24 | 74 | 49
  SARS-CoV-2 DB His-50 at Month 0-Total | 49 | 138 | 22 | 70 | 47
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 33 | 22
  SARS-CoV-2 DB His-50 at Month 0-USA | 25 | 83 | 6 | 29 | 20
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 25 | 44 | 17 | 31 | 20
  SARS-CoV-2 DB His-50 at Month 2-Peru | 22 | 41 | 15 | 31 | 20
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 49 | 115 | 21 | 55 | 35
  SARS-CoV-2 DB His-50 at Month 2-Total | 39 | 106 | 19 | 51 | 32
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 24 | 71 | 4 | 24 | 15
  SARS-CoV-2 DB His-50 at Month 2-USA | 17 | 65 | 4 | 20 | 12
  SARS-CoV-2 DB His-50 at Month 4-Peru: number analyzed (Participants) | 26 | 36 | 16 | 22 | 14
  SARS-CoV-2 DB His-50 at Month 4-Peru | 24 | 31 | 14 | 22 | 14
  SARS-CoV-2 DB His-50 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 40 | 25
  SARS-CoV-2 DB His-50 at Month 4-Total | 31 | 70 | 16 | 37 | 23
  SARS-CoV-2 DB His-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 18 | 11
  SARS-CoV-2 DB His-50 at Month 4-USA | 7 | 39 | 2 | 15 | 9
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 28 | 60 | 18 | 41 | 27
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 24 | 55 | 16 | 41 | 27
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 73 | 147 | 24 | 74 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 50 | 137 | 21 | 69 | 47
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 45 | 87 | 6 | 33 | 22
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 26 | 82 | 5 | 28 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 25 | 45 | 17 | 29 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 22 | 40 | 15 | 29 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 47 | 115 | 21 | 52 | 34
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 38 | 103 | 19 | 48 | 31
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 22 | 70 | 4 | 23 | 14
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 16 | 63 | 4 | 19 | 11
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Peru: number analyzed (Participants) | 26 | 34 | 16 | 20 | 12
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Peru | 22 | 30 | 14 | 20 | 12
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total: number analyzed (Participants) | 38 | 75 | 18 | 37 | 22
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total | 29 | 65 | 16 | 34 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-USA: number analyzed (Participants) | 12 | 41 | 2 | 17 | 10
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-USA | 7 | 35 | 2 | 14 | 8
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 18 | 44 | 14 | 38 | 26
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 15 | 43 | 14 | 38 | 26
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 49 | 96 | 18 | 58 | 43
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 33 | 95 | 18 | 56 | 42
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 31 | 52 | 4 | 20 | 17
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 18 | 52 | 4 | 18 | 16
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 25 | 46 | 16 | 31 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 22 | 42 | 14 | 31 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 49 | 116 | 20 | 55 | 35
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 40 | 107 | 18 | 51 | 33
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 24 | 70 | 4 | 24 | 15
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 18 | 65 | 4 | 20 | 13
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Peru: number analyzed (Participants) | 26 | 37 | 16 | 21 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Peru | 24 | 33 | 14 | 21 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 39 | 25
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total | 32 | 73 | 16 | 36 | 24
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 18 | 11
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-USA | 8 | 40 | 2 | 15 | 10
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 26 | 59 | 17 | 40 | 27
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 22 | 56 | 15 | 40 | 27
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 70 | 143 | 23 | 73 | 49
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 46 | 136 | 21 | 68 | 46
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 44 | 84 | 6 | 33 | 22
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 24 | 80 | 6 | 28 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 25 | 47 | 17 | 31 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 22 | 43 | 15 | 31 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 49 | 117 | 21 | 55 | 35
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 40 | 107 | 19 | 51 | 32
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 24 | 70 | 4 | 24 | 15
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 18 | 64 | 4 | 20 | 12
  SARS-CoV-2 S1 C His-50 at Month 4-Peru: number analyzed (Participants) | 26 | 36 | 16 | 22 | 14
  SARS-CoV-2 S1 C His-50 at Month 4-Peru | 24 | 31 | 14 | 22 | 14
  SARS-CoV-2 S1 C His-50 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 40 | 25
  SARS-CoV-2 S1 C His-50 at Month 4-Total | 32 | 70 | 16 | 37 | 23
  SARS-CoV-2 S1 C His-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 18 | 11
  SARS-CoV-2 S1 C His-50 at Month 4-USA | 8 | 39 | 2 | 15 | 9
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 27 | 60 | 18 | 41 | 27
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 24 | 55 | 16 | 41 | 27
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 71 | 148 | 24 | 73 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 54 | 138 | 22 | 70 | 47
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 32 | 22
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 30 | 83 | 6 | 29 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 23 | 46 | 16 | 30 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 21 | 43 | 14 | 30 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 43 | 115 | 20 | 52 | 35
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 36 | 108 | 18 | 50 | 34
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 20 | 69 | 4 | 22 | 15
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 15 | 65 | 4 | 20 | 14
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Peru: number analyzed (Participants) | 26 | 32 | 15 | 21 | 12
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Peru | 25 | 29 | 13 | 21 | 12
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 38 | 72 | 17 | 39 | 22
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total | 34 | 66 | 15 | 37 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-USA: number analyzed (Participants) | 12 | 40 | 2 | 18 | 10
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-USA | 9 | 37 | 2 | 16 | 8
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 26
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 25 | 58 | 16 | 41 | 26
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 73 | 150 | 24 | 74 | 48
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 53 | 141 | 22 | 69 | 47
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 33 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 28 | 83 | 6 | 28 | 21
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 25 | 46 | 17 | 31 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 22 | 42 | 15 | 31 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 49 | 117 | 21 | 55 | 35
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 40 | 108 | 19 | 52 | 34
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 24 | 71 | 4 | 24 | 15
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 18 | 66 | 4 | 21 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Peru: number analyzed (Participants) | 26 | 37 | 16 | 22 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Peru | 24 | 33 | 14 | 22 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 41 | 25
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total | 32 | 73 | 16 | 38 | 24
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 19 | 11
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-USA | 8 | 40 | 2 | 16 | 10
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 18 | 45 | 14 | 39 | 26
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 15 | 44 | 14 | 39 | 26
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 49 | 99 | 18 | 59 | 43
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 35 | 96 | 18 | 57 | 41
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 31 | 54 | 4 | 20 | 17
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 20 | 52 | 4 | 18 | 15
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 25 | 46 | 16 | 31 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 22 | 42 | 14 | 31 | 20
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 48 | 114 | 20 | 53 | 34
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 38 | 103 | 18 | 50 | 32
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 23 | 68 | 4 | 22 | 14
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 16 | 61 | 4 | 19 | 12
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Peru: number analyzed (Participants) | 26 | 37 | 16 | 22 | 14
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Peru | 24 | 34 | 14 | 22 | 14
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 40 | 25
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total | 32 | 72 | 16 | 37 | 23
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-USA: number analyzed (Participants) | 12 | 43 | 2 | 18 | 11
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-USA | 8 | 38 | 2 | 15 | 9

17. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG1) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2, 4
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
MFI
  2019-nCoV S/293F-1000 at Month 0-Total: number analyzed (Participants) | 53 | 106 | 19 | 62 | 44
  2019-nCoV S/293F-1000 at Month 0-Total | 5989.2 [90.5 to 11296.8] | 11935.2 [4328.6 to 22000] | 22000 [16117.8 to 22000] | 22000 [22000 to 22000] | 22000 [16040.6 to 22000]
  2019-nCoV S/293F-1000 at Month 2-Total: number analyzed (Participants) | 47 | 114 | 21 | 55 | 35
  2019-nCoV S/293F-1000 at Month 2-Total | 2149 [892.8 to 5544.1] | 6736.9 [2053.1 to 14929.9] | 16940.5 [7339 to 22000] | 19418 [9154 to 22000] | 15764.8 [10970.8 to 22000]
  2019-nCoV S/293F-1000 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 41 | 25
  2019-nCoV S/293F-1000 at Month 4-Total | 1159.1 [469.4 to 2136.5] | 2032.6 [957.7 to 8274.9] | 7015.6 [2425.8 to 15008.7] | 11395.5 [4827 to 19747.2] | 13465.2 [5921.2 to 20349.3]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 50 | 92 | 16 | 59 | 43
  229E-RBD-50 at Month 0-Total | 4100.9 [1900.8 to 7294.5] | 5351.8 [3432.4 to 8184.1] | 6758.9 [3951.3 to 8605] | 7487.5 [4141 to 9716] | 5035.8 [3682 to 6589.4]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 49 | 114 | 16 | 48 | 34
  229E-RBD-50 at Month 2-Total | 4701.2 [2838.5 to 6825.5] | 4798 [2842.5 to 7790.1] | 7490.1 [4311.1 to 8744.1] | 5405.2 [3093.4 to 8470.2] | 5567.6 [4189.1 to 7235.9]
  229E-RBD-50 at Month 4-Total: number analyzed (Participants) | 38 | 72 | 16 | 35 | 20
  229E-RBD-50 at Month 4-Total | 5162.5 [3855.9 to 7221.9] | 6192.8 [3392 to 9030.2] | 8425.6 [6552.2 to 10927.2] | 7296.2 [5270.8 to 9552.1] | 6106.1 [5264.1 to 8204.1]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 144 | 18 | 60 | 46
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 14002.2 [6702.2 to 21425.9] | 14944.4 [9753.9 to 22000] | 18253.1 [12441.3 to 21369.4] | 13857.6 [7431 to 21445.4] | 10321.2 [5614.9 to 15196.4]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 48 | 115 | 16 | 50 | 34
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 10239.5 [7166.4 to 18628.6] | 9586.8 [6383.6 to 15287.4] | 15170.5 [9241.1 to 18084.6] | 8577.8 [5176.2 to 14077.9] | 6796.5 [4171.5 to 12932.1]
  HCoV-229E S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 38 | 78 | 18 | 37 | 23
  HCoV-229E S1S2 ECD His-50 at Month 4-Total | 10870.5 [6480.4 to 17301.9] | 9447.5 [6667.2 to 14856.6] | 11755.5 [8332.2 to 14752.1] | 9325.8 [5152.5 to 14824] | 9645.5 [4611 to 13284.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 144 | 17 | 60 | 46
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 11218.4 [4227.2 to 17991.8] | 15650.4 [10267.8 to 22000] | 18108.8 [7185 to 20531] | 17008.2 [10572.9 to 22000] | 14307.9 [7145.9 to 21912.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 49 | 114 | 16 | 49 | 35
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 12434.8 [7962.8 to 18575.8] | 12646.1 [7867.9 to 19532.1] | 14461.6 [7353.3 to 21226.6] | 16030 [6863 to 22000] | 14744.2 [9894.9 to 20172.4]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 39 | 25
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total | 9754 [5536.6 to 18087.8] | 13201.2 [6891.8 to 20931.6] | 15596.3 [8533.3 to 19332.8] | 16039.8 [9555.5 to 22000] | 12057.8 [7646.8 to 18609.8]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 143 | 18 | 61 | 46
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 1328.1 [740.6 to 2715.1] | 1890.5 [421 to 3400.5] | 787.2 [1 to 2116.8] | 128.8 [1 to 2817.5] | 384.8 [1 to 1827.5]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 39 | 111 | 15 | 49 | 25
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 2430 [1111.6 to 4146.8] | 2124.8 [887.6 to 4072.9] | 1430 [125.5 to 3789.6] | 863 [1 to 3723.5] | 196 [1 to 1349.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 17 | 37 | 23
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total | 1370.5 [793.9 to 2813.2] | 1990.5 [791.8 to 3077.6] | 1411 [866.5 to 1976.8] | 1123 [497.8 to 3821.2] | 947.2 [326.8 to 2567.6]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 144 | 18 | 60 | 46
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 21718.6 [11765.6 to 22000] | 22000 [17471.2 to 22000] | 20677.4 [15975 to 22000] | 21907.4 [19535 to 22000] | 22000 [17563.7 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 49 | 115 | 16 | 50 | 34
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 22000 [14469.5 to 22000] | 22000 [14622.4 to 22000] | 21644.5 [12189.4 to 22000] | 22000 [16390.9 to 22000] | 22000 [18397.4 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 38 | 24
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total | 18483.5 [10544.5 to 22000] | 22000 [13327.5 to 22000] | 21513.2 [13513.9 to 22000] | 22000 [17186.5 to 22000] | 22000 [16949.7 to 22000]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 51 | 97 | 16 | 56 | 42
  HKU1-RBD-50 at Month 0-Total | 3326.8 [955.4 to 4966.1] | 4487.5 [2979.8 to 6232] | 5480.8 [3668.6 to 7159.3] | 5309.2 [3624.6 to 8638.2] | 3714.6 [2070.3 to 5822.9]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 47 | 112 | 16 | 47 | 34
  HKU1-RBD-50 at Month 2-Total | 3843 [2609.4 to 5512.5] | 3835.9 [1945.1 to 5303.4] | 5927.4 [3782.1 to 8082.2] | 4881.2 [1952.2 to 7723] | 3902.6 [1972.3 to 5690.3]
  HKU1-RBD-50 at Month 4-Total: number analyzed (Participants) | 37 | 68 | 16 | 34 | 21
  HKU1-RBD-50 at Month 4-Total | 3976.5 [2390 to 7096.8] | 4933.5 [2869.3 to 7746.8] | 7185.2 [4821.9 to 12208.1] | 6354.1 [4134.8 to 8926.9] | 5575.8 [3624 to 6671]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 51 | 96 | 16 | 58 | 42
  NL63-RBD-50 at Month 0-Total | 11577 [9062.4 to 15938.8] | 12831.8 [9340 to 16679.6] | 10709.4 [8215.4 to 13102.1] | 12869.4 [8782.1 to 16942.2] | 10772.1 [7934.6 to 13885.8]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 49 | 115 | 16 | 51 | 34
  NL63-RBD-50 at Month 2-Total | 15942.5 [13683.2 to 20130.5] | 14045 [10306.9 to 17711.2] | 16062.2 [11906.2 to 20001.2] | 13088.2 [8506.8 to 19241.6] | 11879.5 [8520.2 to 15218.8]
  NL63-RBD-50 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 39 | 25
  NL63-RBD-50 at Month 4-Total | 16414.2 [14140.4 to 19850] | 16559.2 [12559.5 to 19641.5] | 17690.1 [15662.1 to 21231.3] | 15559.8 [11989.5 to 20530.5] | 15900.2 [12375.8 to 18128.8]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 51 | 96 | 16 | 55 | 42
  OC43-RBD-50 at Month 0-Total | 3364.8 [1423.4 to 5812.4] | 4057.5 [2340.8 to 6578.6] | 3836.9 [2239.9 to 6492.2] | 4979.5 [3344.9 to 8658] | 3653.9 [2134.6 to 6225]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 49 | 114 | 15 | 47 | 34
  OC43-RBD-50 at Month 2-Total | 4004.2 [2449 to 8214] | 4138.5 [2234.2 to 6051.5] | 6048 [2454.2 to 9758.5] | 4726.5 [2750 to 9097.6] | 4209.2 [2684 to 6779.2]
  OC43-RBD-50 at Month 4-Total: number analyzed (Participants) | 37 | 72 | 15 | 35 | 22
  OC43-RBD-50 at Month 4-Total | 3639.8 [2183.8 to 5068.2] | 4952.2 [2098.1 to 7392.9] | 6118 [4052.6 to 9482.8] | 7069.8 [5100.8 to 10583.5] | 6074.8 [3952.9 to 9225]
  SARS-CoV-2 DB His-1000 at Month 0-Total: number analyzed (Participants) | 72 | 148 | 24 | 74 | 49
  SARS-CoV-2 DB His-1000 at Month 0-Total | 1172.4 [4.9 to 3036.6] | 3808 [949.2 to 10571] | 13049.5 [7157.2 to 22000] | 20453.6 [6304.2 to 22000] | 15945.2 [5574.2 to 22000]
  SARS-CoV-2 DB His-1000 at Month 2-Total: number analyzed (Participants) | 49 | 115 | 21 | 55 | 35
  SARS-CoV-2 DB His-1000 at Month 2-Total | 676.2 [196.5 to 1679.2] | 1196 [348.6 to 3746.6] | 5149 [1728.2 to 10064] | 5809 [1712.8 to 15047.1] | 4720 [2789.8 to 11054.6]
  SARS-CoV-2 DB His-1000 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 40 | 25
  SARS-CoV-2 DB His-1000 at Month 4-Total | 363.6 [192.8 to 658.4] | 526.5 [222.4 to 2206.1] | 1479.2 [453.1 to 4343] | 2783 [1316.9 to 7014.1] | 3621 [1590 to 5098]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total: number analyzed (Participants) | 73 | 147 | 24 | 74 | 49
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total | 1591.8 [113 to 4922.2] | 10582 [2114.2 to 22000] | 22000 [11571.4 to 22000] | 22000 [14010.6 to 22000] | 16037.8 [3105 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total: number analyzed (Participants) | 47 | 115 | 21 | 52 | 34
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total | 614.8 [287.9 to 1356] | 1910.8 [554.2 to 5501.4] | 6201.5 [2773.5 to 13504.8] | 6099.5 [2365.7 to 12367.8] | 4573.9 [1131.8 to 8607.4]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total: number analyzed (Participants) | 38 | 75 | 18 | 37 | 22
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total | 218.9 [135.8 to 434.1] | 465 [237.4 to 1591.2] | 1442.9 [233.9 to 3319.8] | 1442.5 [452.5 to 4576.2] | 801.5 [432.8 to 1695.3]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total: number analyzed (Participants) | 49 | 96 | 18 | 58 | 43
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total | 838.5 [1 to 1488.5] | 3318.9 [1198 to 8993.9] | 13555.6 [8042.8 to 20075] | 15429.4 [9351.4 to 22000] | 14558.5 [3989.8 to 22000]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total: number analyzed (Participants) | 49 | 116 | 20 | 55 | 35
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total | 434.8 [211.5 to 1337.2] | 1093.4 [401.2 to 3314.4] | 4634.2 [1322.6 to 10511] | 6504.2 [1883.8 to 11889.5] | 4875 [2939.5 to 12514.6]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 39 | 25
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total | 292 [151.3 to 487.3] | 436.5 [239.4 to 1852.6] | 1634.2 [382.5 to 4709.4] | 2848 [1081.5 to 6415.8] | 3884.2 [1477.5 to 6633.2]
  SARS-CoV-2 S1 C His-1000 at Month 0-Total: number analyzed (Participants) | 70 | 143 | 23 | 73 | 49
  SARS-CoV-2 S1 C His-1000 at Month 0-Total | 837.1 [53.6 to 2356.2] | 3224.8 [566.9 to 8992.8] | 11397 [5598.4 to 22000] | 20747.2 [6541.8 to 22000] | 18275.8 [7261 to 22000]
  SARS-CoV-2 S1 C His-1000 at Month 2-Total: number analyzed (Participants) | 49 | 117 | 21 | 55 | 35
  SARS-CoV-2 S1 C His-1000 at Month 2-Total | 375.5 [156.8 to 1260.5] | 879.5 [226.8 to 3227] | 3926.5 [1530.8 to 12636] | 5654.2 [1635.5 to 16795.2] | 4787.5 [2606.9 to 13220]
  SARS-CoV-2 S1 C His-1000 at Month 4-Total: number analyzed (Participants) | 38 | 79 | 18 | 40 | 25
  SARS-CoV-2 S1 C His-1000 at Month 4-Total | 228 [124.6 to 463.1] | 383.8 [193.2 to 2039.6] | 1493.2 [418.3 to 5506.1] | 2603.9 [1040 to 7404.1] | 3391.8 [1766.5 to 6985.5]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total: number analyzed (Participants) | 71 | 148 | 24 | 73 | 49
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total | 839.2 [62.8 to 3136.2] | 3872.8 [1031.1 to 10614.9] | 10200 [3868.4 to 18939.6] | 15822 [9604.5 to 22000] | 14078.2 [9060 to 18504]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total: number analyzed (Participants) | 43 | 115 | 20 | 52 | 35
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total | 402 [169.1 to 1450.5] | 1496.5 [355.8 to 4277.1] | 6103.8 [1693.4 to 10371.4] | 6823.5 [2420.5 to 14742.1] | 8218.5 [2871.2 to 12878.6]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total: number analyzed (Participants) | 38 | 72 | 17 | 39 | 22
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total | 290.8 [179.1 to 690] | 710.2 [164.7 to 2857.7] | 1147 [463.2 to 4076.8] | 3203.2 [1156.2 to 7891.5] | 4619.9 [1360 to 7799]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total: number analyzed (Participants) | 73 | 150 | 24 | 74 | 48
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total | 4511.2 [182 to 9507.8] | 10463.4 [4513.8 to 21974.2] | 21026.6 [14574.4 to 22000] | 22000 [19015.4 to 22000] | 22000 [18083.9 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total: number analyzed (Participants) | 49 | 117 | 21 | 55 | 35
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total | 2497.5 [1173 to 5380.2] | 5993.8 [2335.8 to 12505.5] | 16653.5 [5921.5 to 22000] | 17261.2 [8244.2 to 22000] | 17681.8 [9882 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 41 | 25
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total | 1456.8 [642.3 to 2659.9] | 2203.4 [1047.7 to 8793.9] | 7099.9 [2271.6 to 13897.5] | 11311.2 [5053 to 18428.2] | 11779.2 [5739 to 19179.8]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total: number analyzed (Participants) | 49 | 99 | 18 | 59 | 43
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total | 325.8 [1 to 1308.5] | 2031.2 [326.8 to 10576.4] | 5595.2 [3346 to 22000] | 22000 [9695.6 to 22000] | 15796.8 [4864.1 to 22000]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total: number analyzed (Participants) | 48 | 114 | 20 | 53 | 34
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total | 99.6 [9.4 to 405.8] | 472 [46.9 to 2230.9] | 3360.2 [538 to 14750.2] | 4301 [1118.8 to 11382.8] | 3229.6 [1033.2 to 11824.9]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total: number analyzed (Participants) | 38 | 80 | 18 | 40 | 25
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total | 44.4 [18.7 to 145.8] | 165 [19.1 to 581.1] | 583.4 [92.5 to 3312.4] | 1914.2 [403.9 to 4041.2] | 1798.5 [515.5 to 4191.5]

18. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG3) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 29 | 59 | 18 | 41 | 28
  2019-nCoV S/293F-50 at Month 0-Peru | 25 | 54 | 17 | 41 | 28
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 74 | 147 | 24 | 74 | 50
  2019-nCoV S/293F-50 at Month 0-Total | 52 | 136 | 23 | 71 | 48
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 33 | 22
  2019-nCoV S/293F-50 at Month 0-USA | 27 | 82 | 6 | 30 | 20
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  2019-nCoV S/293F-50 at Month 2-Peru | 0 | 11 | 6 | 7 | 2
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  2019-nCoV S/293F-50 at Month 2-Total | 4 | 50 | 7 | 16 | 6
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  2019-nCoV S/293F-50 at Month 2-USA | 4 | 39 | 1 | 9 | 4
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 28 | 60 | 18 | 41 | 28
  SARS-CoV-2 DB His-50 at Month 0-Peru | 24 | 48 | 15 | 41 | 26
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 73 | 148 | 24 | 74 | 50
  SARS-CoV-2 DB His-50 at Month 0-Total | 42 | 117 | 21 | 70 | 45
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 33 | 22
  SARS-CoV-2 DB His-50 at Month 0-USA | 18 | 69 | 6 | 29 | 19
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 DB His-50 at Month 2-Peru | 0 | 4 | 4 | 4 | 2
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 DB His-50 at Month 2-Total | 2 | 23 | 5 | 10 | 5
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 DB His-50 at Month 2-USA | 2 | 19 | 1 | 6 | 3
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 60 | 18 | 41 | 28
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 26 | 55 | 16 | 41 | 28
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 73 | 148 | 24 | 74 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 56 | 138 | 22 | 71 | 48
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 33 | 22
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 30 | 83 | 6 | 30 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 0 | 8 | 6 | 6 | 2
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 4 | 46 | 7 | 13 | 6
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 4 | 38 | 1 | 7 | 4
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 28 | 59 | 18 | 41 | 28
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 23 | 51 | 16 | 40 | 28
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 72 | 147 | 24 | 74 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 39 | 126 | 22 | 68 | 48
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 33 | 22
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 16 | 75 | 6 | 28 | 20
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 0 | 6 | 4 | 6 | 2
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 3 | 29 | 5 | 14 | 6
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 3 | 23 | 1 | 8 | 4
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 25 | 50 | 16 | 40 | 28
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 74 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 45 | 123 | 22 | 69 | 48
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 33 | 22
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 20 | 73 | 6 | 29 | 20
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 0 | 6 | 5 | 6 | 2
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 3 | 31 | 6 | 14 | 6
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 3 | 25 | 1 | 8 | 4
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 26 | 54 | 16 | 41 | 28
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 72 | 148 | 24 | 74 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 55 | 136 | 22 | 72 | 48
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 43 | 87 | 6 | 33 | 22
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 29 | 82 | 6 | 31 | 20
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 0 | 12 | 7 | 8 | 2
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 4 | 55 | 8 | 16 | 6
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 4 | 43 | 1 | 8 | 4
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 25 | 56 | 17 | 41 | 28
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 74 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 51 | 138 | 23 | 71 | 48
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 33 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 26 | 82 | 6 | 30 | 20
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 0 | 9 | 7 | 7 | 2
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 4 | 46 | 8 | 16 | 6
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 4 | 37 | 1 | 9 | 4
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 29 | 60 | 18 | 41 | 28
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 25 | 51 | 16 | 41 | 28
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 74 | 148 | 24 | 74 | 50
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 45 | 127 | 22 | 69 | 47
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 33 | 22
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 20 | 76 | 6 | 28 | 19
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 0 | 10 | 6 | 7 | 2
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 4 | 44 | 7 | 15 | 6
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 4 | 34 | 1 | 8 | 4

19. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG3) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
MFI
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 74 | 147 | 24 | 74 | 50
  2019-nCoV S/293F-50 at Month 0-Total | 2775.6 [226.4 to 7398.3] | 5366.5 [3056.1 to 9837.5] | 5835.1 [3507.9 to 10801.1] | 11878.2 [7048.9 to 17857.1] | 10388.5 [5691.6 to 18870.2]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  2019-nCoV S/293F-50 at Month 2-Total | 3573.2 [3027 to 5723.6] | 2217.9 [628.8 to 4404.2] | 2597 [738.2 to 3307] | 3720.4 [2910.6 to 5906.6] | 3562 [2814.6 to 5474.5]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 68 | 148 | 24 | 71 | 47
  229E-RBD-50 at Month 0-Total | 131 [1 to 377.5] | 235.2 [82.4 to 474.7] | 143 [29.7 to 254.1] | 329 [75.9 to 626.8] | 374 [1 to 660.9]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 61 | 9 | 18 | 7
  229E-RBD-50 at Month 2-Total | 8.9 [1 to 24.3] | 1 [1 to 61.8] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 10.4]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 72 | 50
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 32 [1 to 127.2] | 29.2 [1 to 136.5] | 7.6 [1 to 57.2] | 1 [1 to 51.9] | 1 [1 to 17.9]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 388.8 [110.7 to 1489.3] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 15.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 73 | 149 | 23 | 73 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 268.2 [66.5 to 718.8] | 459.5 [163 to 1213.2] | 328.5 [196.2 to 776.4] | 518.8 [176 to 1390.2] | 383 [1 to 1697.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 626.8 [341.8 to 2818.4] | 189.6 [1 to 714.8] | 142.2 [1 to 318.2] | 97.2 [1 to 416.1] | 562.2 [160.1 to 1378.8]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 72 | 50
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 7.1 [1 to 54.1] | 9.8 [1 to 69.5] | 1 [1 to 33.4] | 1 [1 to 54.1] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 15.4 [1 to 958.1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 73 | 149 | 24 | 73 | 49
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 562.8 [158.8 to 1637] | 611.5 [164.2 to 2449] | 424.5 [100.9 to 943.8] | 485.2 [132 to 1650.5] | 131 [1 to 1264.2]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 61 | 9 | 18 | 6
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 802.8 [565.2 to 6271] | 10.2 [1 to 570] | 1 [1 to 32.2] | 1 [1 to 255.2] | 371.1 [56.4 to 1543.3]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 72 | 145 | 24 | 73 | 48
  HKU1-RBD-50 at Month 0-Total | 122.6 [1 to 328.4] | 196.8 [97.5 to 312.8] | 132.9 [37.5 to 254.9] | 250.8 [59.8 to 446.8] | 270.8 [1 to 546.2]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HKU1-RBD-50 at Month 2-Total | 66.4 [1 to 149.8] | 1 [1 to 1.9] | 1 [1 to 1] | 1 [1 to 167.2] | 1 [1 to 59.1]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 67 | 141 | 22 | 67 | 49
  NL63-RBD-50 at Month 0-Total | 191.5 [1 to 386.4] | 215.2 [35.2 to 453] | 206.6 [70.1 to 400.2] | 275.5 [74.5 to 518.4] | 195.8 [1 to 439.5]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  NL63-RBD-50 at Month 2-Total | 61.8 [1 to 130] | 1 [1 to 37.7] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 41.4]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 71 | 148 | 24 | 71 | 50
  OC43-RBD-50 at Month 0-Total | 102.2 [1 to 261.1] | 151.9 [12.1 to 313.6] | 122.9 [1 to 260.3] | 198 [42.6 to 453.5] | 154.1 [1 to 449.1]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  OC43-RBD-50 at Month 2-Total | 2.8 [1 to 16] | 1 [1 to 16.8] | 1 [1 to 1] | 1 [1 to 40.6] | 1 [1 to 29.5]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 73 | 148 | 24 | 74 | 50
  SARS-CoV-2 DB His-50 at Month 0-Total | 549 [61.5 to 1848.5] | 1472.5 [570.2 to 2942.9] | 1848.9 [796.4 to 3564.9] | 3532.5 [1978.6 to 5226.4] | 3818.5 [1378.9 to 5591.2]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 DB His-50 at Month 2-Total | 430.4 [338.2 to 734.1] | 111.8 [1 to 790.6] | 494.2 [19.5 to 897.5] | 691.5 [9.6 to 1343.6] | 655.5 [248.9 to 1001.5]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 73 | 148 | 24 | 74 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 3858.8 [408.8 to 8570.2] | 6125 [3010 to 11582.6] | 8722.4 [4573.3 to 12243.4] | 13805.6 [6730.1 to 20791.1] | 11790.8 [4678.7 to 18578.9]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 4270.1 [1334.9 to 7545.8] | 1596.1 [308.2 to 3591.9] | 726.5 [521 to 1330.8] | 2358.2 [583.1 to 4394.3] | 3132.5 [1966.4 to 4286.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 72 | 147 | 24 | 74 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 466.6 [55.1 to 1777.4] | 1235.5 [474.1 to 2423] | 1634.1 [1044.4 to 3244.7] | 4180.4 [2199.1 to 6351.9] | 4158.9 [1424.2 to 6264.8]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 551 [402.3 to 655.2] | 178.6 [1 to 991.2] | 241.2 [101.5 to 1153] | 681.2 [276.2 to 1079.2] | 966.2 [755.1 to 1617.6]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 74 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 542.2 [83.8 to 1428.8] | 1394.8 [354 to 2617.2] | 1690.2 [870.9 to 3543.7] | 4453.4 [2463.8 to 6519.8] | 4152.1 [2270.4 to 7842.4]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 421.1 [271.6 to 737.2] | 222.4 [18.9 to 1120.9] | 781.2 [28 to 1880] | 1168.6 [377 to 1630.4] | 1200.5 [768 to 1534.6]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 72 | 148 | 24 | 74 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 4162.8 [799.6 to 10622.6] | 6037.8 [3290.1 to 14853.2] | 7290.6 [5033 to 17937.1] | 15804.8 [7974.9 to 22000] | 15218.4 [8344.4 to 22000]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 6799.9 [2662.2 to 13522] | 3986.6 [1958.4 to 9672.4] | 2566.2 [1660.2 to 5027.2] | 5121.6 [2066.5 to 10043.6] | 8445.8 [5726.5 to 17144.9]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 74 | 149 | 24 | 74 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 2129 [311.9 to 4773.1] | 3914.5 [2186.5 to 6376.5] | 3562.6 [2272.2 to 6921.2] | 8685.9 [5554.5 to 11434.8] | 7397.4 [4187.8 to 13306.2]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 2365.4 [2072.2 to 2947] | 1729.8 [403.1 to 2896.8] | 1699.2 [539 to 2524.5] | 2640.1 [1741.9 to 3770.8] | 2402.2 [2008 to 3440.5]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 74 | 148 | 24 | 74 | 50
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 430.8 [2.9 to 2020.1] | 1814.2 [314.4 to 5209.5] | 3141.2 [1434.1 to 8485.8] | 7721.8 [3836 to 11832.4] | 5454 [2733.5 to 11251.8]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 326.8 [245.1 to 666.6] | 234.8 [6.5 to 1381.2] | 903 [144.8 to 1502.8] | 997.2 [562.6 to 1721] | 1713 [749.8 to 1865.8]

20. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgA) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  2019-nCoV S/293F-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  2019-nCoV S/293F-50 at Month 0-Peru | 25 | 57 | 16 | 41 | 28
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  2019-nCoV S/293F-50 at Month 0-Total | 53 | 137 | 22 | 70 | 47
  2019-nCoV S/293F-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  2019-nCoV S/293F-50 at Month 0-USA | 28 | 80 | 6 | 29 | 19
  2019-nCoV S/293F-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  2019-nCoV S/293F-50 at Month 2-Peru | 0 | 11 | 7 | 8 | 2
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  2019-nCoV S/293F-50 at Month 2-Total | 4 | 52 | 8 | 16 | 6
  2019-nCoV S/293F-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  2019-nCoV S/293F-50 at Month 2-USA | 4 | 41 | 1 | 8 | 4
  SARS-CoV-2 DB His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 DB His-50 at Month 0-Peru | 21 | 51 | 16 | 41 | 28
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 DB His-50 at Month 0-Total | 41 | 109 | 22 | 66 | 45
  SARS-CoV-2 DB His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 DB His-50 at Month 0-USA | 20 | 58 | 6 | 25 | 17
  SARS-CoV-2 DB His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 DB His-50 at Month 2-Peru | 0 | 8 | 6 | 7 | 2
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 DB His-50 at Month 2-Total | 3 | 37 | 7 | 12 | 6
  SARS-CoV-2 DB His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 DB His-50 at Month 2-USA | 3 | 29 | 1 | 5 | 4
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Peru | 26 | 54 | 18 | 39 | 27
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 56 | 127 | 24 | 68 | 47
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-USA | 30 | 73 | 6 | 29 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Peru | 0 | 12 | 8 | 8 | 2
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 3 | 47 | 9 | 14 | 6
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-USA | 3 | 35 | 1 | 6 | 4
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Peru | 26 | 58 | 16 | 41 | 28
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 54 | 140 | 22 | 70 | 47
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-USA | 28 | 82 | 6 | 29 | 19
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Peru | 0 | 13 | 7 | 8 | 2
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 4 | 55 | 8 | 15 | 6
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-USA | 4 | 42 | 1 | 7 | 4
  SARS-CoV-2 S1 C His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 S1 C His-50 at Month 0-Peru | 26 | 55 | 16 | 41 | 28
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 51 | 132 | 22 | 70 | 47
  SARS-CoV-2 S1 C His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 S1 C His-50 at Month 0-USA | 25 | 77 | 6 | 29 | 19
  SARS-CoV-2 S1 C His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S1 C His-50 at Month 2-Peru | 0 | 10 | 7 | 8 | 2
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 4 | 48 | 8 | 15 | 6
  SARS-CoV-2 S1 C His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S1 C His-50 at Month 2-USA | 4 | 38 | 1 | 7 | 4
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Peru | 5 | 32 | 12 | 33 | 25
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 11 | 54 | 15 | 51 | 37
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-USA | 6 | 22 | 3 | 18 | 12
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Peru | 0 | 3 | 2 | 5 | 1
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 1 | 16 | 3 | 7 | 4
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-USA | 1 | 13 | 1 | 2 | 3
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru: number analyzed (Participants) | 29 | 62 | 18 | 41 | 28
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Peru | 25 | 53 | 16 | 41 | 28
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 51 | 127 | 22 | 68 | 47
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA: number analyzed (Participants) | 45 | 88 | 6 | 34 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-USA | 26 | 74 | 6 | 27 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Peru | 0 | 8 | 6 | 8 | 2
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 4 | 47 | 7 | 15 | 6
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-USA | 4 | 39 | 1 | 7 | 4
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru: number analyzed (Participants) | 23 | 46 | 11 | 35 | 25
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Peru | 17 | 37 | 10 | 35 | 25
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 64 | 91 | 15 | 62 | 43
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 31 | 66 | 14 | 57 | 39
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA: number analyzed (Participants) | 41 | 45 | 4 | 27 | 18
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-USA | 14 | 29 | 4 | 22 | 14
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru: number analyzed (Participants) | 0 | 16 | 8 | 8 | 2
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Peru | 0 | 7 | 6 | 8 | 2
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 1 | 33 | 7 | 14 | 5
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA: number analyzed (Participants) | 4 | 46 | 1 | 10 | 5
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-USA | 1 | 26 | 1 | 6 | 3

21. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgA) by Region and COVID-19 Severity Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
MFI
  2019-nCoV S/293F-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  2019-nCoV S/293F-250 at Month 0-Total | 712.6 [84.3 to 2433.4] | 1591.4 [535.4 to 4673.6] | 6170 [2483.8 to 10780.6] | 3396.5 [2324.1 to 9464.5] | 3914.4 [2241.7 to 6653.8]
  2019-nCoV S/293F-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  2019-nCoV S/293F-250 at Month 2-Total | 2994.4 [1566.1 to 4154.5] | 650.6 [368.1 to 1486.9] | 2644.8 [1731.2 to 3965] | 1280.2 [402.6 to 2513.9] | 2037.5 [1812.9 to 4390.5]
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  2019-nCoV S/293F-50 at Month 0-Total | 3018.9 [355.2 to 7725.2] | 5220.1 [2267.2 to 11085.5] | 13988.5 [7764.6 to 22000] | 10462 [5808.1 to 20569.1] | 11893.9 [7800.2 to 15405.3]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  2019-nCoV S/293F-50 at Month 2-Total | 8806.4 [5425.2 to 11275.7] | 2630 [1486 to 4731.1] | 7052 [5451.2 to 9517.5] | 4473.9 [1626.4 to 7328.2] | 6588 [6082.8 to 11702.9]
  229E-RBD-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  229E-RBD-250 at Month 0-Total | 104 [73.2 to 190.6] | 115 [57.6 to 214.9] | 173.2 [103.1 to 303.9] | 170.5 [111.9 to 342.6] | 162.8 [97.8 to 317.1]
  229E-RBD-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  229E-RBD-250 at Month 2-Total | 84.2 [72.9 to 90.4] | 85.5 [56.6 to 177.2] | 87.8 [72.5 to 209.8] | 129 [60.3 to 178.8] | 305.2 [99.2 to 451.5]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  229E-RBD-50 at Month 0-Total | 460.8 [300.1 to 766.3] | 443.9 [223.1 to 859.8] | 644.4 [407.9 to 1120.8] | 642.2 [420.2 to 1264.8] | 603.1 [357.1 to 1162.1]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  229E-RBD-50 at Month 2-Total | 332.9 [261.9 to 370.4] | 334.1 [204.4 to 687.4] | 308 [250.2 to 635.5] | 452.1 [238.4 to 704.3] | 938 [300.4 to 1191.2]
  HCoV-229E S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-229E S1S2 ECD His-250 at Month 0-Total | 118 [74.4 to 245.9] | 99.4 [40.8 to 211.4] | 116.4 [64.4 to 217.6] | 135.2 [64.6 to 287] | 107.6 [60.9 to 234.2]
  HCoV-229E S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-229E S1S2 ECD His-250 at Month 2-Total | 95.8 [55.8 to 149.3] | 110.4 [47 to 235.8] | 156.8 [128 to 173.8] | 174.6 [68.5 to 372.7] | 345 [87.2 to 373.8]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 498.9 [294.7 to 977.8] | 408.2 [161.1 to 884.2] | 466.4 [279.6 to 894.1] | 575 [243.9 to 1077.5] | 401.2 [227.3 to 890.9]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 363.5 [228 to 576.5] | 464.9 [163.2 to 891.3] | 585.8 [387 to 713.2] | 681.4 [225.4 to 1414.2] | 913 [261.6 to 1305.5]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 0-Total | 178.6 [114.9 to 431.7] | 320.8 [127.3 to 726.9] | 516.6 [212.5 to 1008.7] | 533 [286.6 to 1169.5] | 482 [165.5 to 1415.3]
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-HKU1 N5 S1S2 ECD His-250 at Month 2-Total | 484.9 [290.8 to 823.1] | 278 [134.6 to 828.6] | 650.8 [251.5 to 907.8] | 362.5 [181.4 to 756.4] | 379.8 [224.9 to 1769]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 744.9 [524.9 to 1694.9] | 1302.8 [560.1 to 2915.9] | 2011.9 [883.1 to 3873.5] | 2137.2 [1164.5 to 4296.5] | 1911.2 [691.1 to 4071.1]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 1952.2 [1178.2 to 3191.1] | 1115.2 [477.5 to 2850.4] | 2676.5 [718 to 4025.5] | 1755 [758.9 to 2820.9] | 1009.5 [718.2 to 5220.2]
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-NL63 S1S2 ECD His-250 at Month 0-Total | 22.5 [10.6 to 46] | 18 [7.6 to 37.1] | 25.1 [11.4 to 66.2] | 32.8 [9.8 to 63.5] | 15.6 [8.1 to 34.3]
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-NL63 S1S2 ECD His-250 at Month 2-Total | 23.1 [16.6 to 34.8] | 21.1 [9.2 to 40.9] | 27 [14.5 to 169] | 20.9 [11.5 to 44.6] | 22.5 [3.2 to 41.4]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 89 [39.5 to 208.1] | 76.6 [31.5 to 162.8] | 96.4 [22.2 to 186.6] | 136.2 [31.1 to 249.8] | 70.5 [25.3 to 133.9]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 5
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 119.8 [78.1 to 173.4] | 85.9 [39.5 to 174.1] | 219.5 [87.8 to 852.5] | 77.6 [55 to 156.6] | 31.8 [1 to 98]
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-OC43 S1S2 ECD His-250 at Month 0-Total | 535.6 [354.1 to 1191.9] | 800.9 [296.2 to 1898.2] | 1031.4 [437.4 to 1811.7] | 1124.2 [534.1 to 2245.1] | 879.1 [354.9 to 2375.8]
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-OC43 S1S2 ECD His-250 at Month 2-Total | 736.9 [633.8 to 928.6] | 745.4 [290.9 to 1811] | 897.2 [713 to 1340.5] | 876.5 [400.8 to 1654.6] | 1083 [377.8 to 3124.8]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 2260 [1354.8 to 4344.1] | 3069.2 [1200.4 to 6140.9] | 3915.4 [1775.8 to 6449.9] | 4348 [2009.9 to 7600.6] | 3272.5 [1648.2 to 7296.4]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 2964.2 [2387.2 to 3715.1] | 2630.5 [1146.8 to 6272] | 3230 [1773.8 to 4732] | 3524.8 [1720.3 to 5816.1] | 2436 [1223 to 8469.6]
  HKU1-RBD-250 at Month 0-Total: number analyzed (Participants) | 73 | 150 | 24 | 75 | 50
  HKU1-RBD-250 at Month 0-Total | 98 [60.8 to 190] | 102 [52.8 to 192.8] | 159.5 [106.3 to 223.6] | 173.8 [107.4 to 328.9] | 132.2 [81.4 to 218.8]
  HKU1-RBD-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HKU1-RBD-250 at Month 2-Total | 87.6 [82 to 386.8] | 88.2 [44.1 to 157.1] | 95.2 [84 to 289.5] | 144.1 [80.7 to 275.6] | 157.2 [120.6 to 271.6]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 73 | 150 | 24 | 75 | 50
  HKU1-RBD-50 at Month 0-Total | 410.5 [269 to 832.5] | 389.2 [224.2 to 736.3] | 589.5 [378.2 to 855.4] | 618.5 [381 to 1212.4] | 445.4 [309.2 to 817.4]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  HKU1-RBD-50 at Month 2-Total | 378.2 [316.6 to 1339.9] | 376.6 [155.5 to 614.6] | 364.8 [333 to 774.5] | 605 [360.1 to 1031.8] | 536.2 [386.9 to 859.6]
  NL63-RBD-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  NL63-RBD-250 at Month 0-Total | 307.4 [178.4 to 592.9] | 276.6 [139.7 to 491.9] | 411 [202.4 to 877.5] | 366 [201.8 to 936.5] | 302.8 [192.6 to 612.1]
  NL63-RBD-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  NL63-RBD-250 at Month 2-Total | 184 [171.3 to 208.7] | 328.1 [152.5 to 530.3] | 374.8 [232.8 to 1210] | 332.6 [139.2 to 937.8] | 226.8 [169.5 to 1207.9]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  NL63-RBD-50 at Month 0-Total | 1208.5 [775.6 to 2311.5] | 1093.5 [584.3 to 2096.1] | 1686 [888 to 3298.7] | 1405.8 [798.8 to 3598] | 1192.4 [842.6 to 2416.2]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  NL63-RBD-50 at Month 2-Total | 743.5 [685.2 to 839.5] | 1279.4 [590 to 2185.1] | 1185.8 [942.5 to 3301.2] | 1183.9 [629.3 to 3318.1] | 869.8 [566.4 to 3704.4]
  OC43-RBD-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  OC43-RBD-250 at Month 0-Total | 126.5 [67.9 to 257.8] | 100.4 [59.4 to 225.1] | 139.1 [78.8 to 257.6] | 168 [84.2 to 326.6] | 143.2 [89.6 to 223.7]
  OC43-RBD-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  OC43-RBD-250 at Month 2-Total | 152.4 [64.4 to 270.4] | 105.2 [57.4 to 258.2] | 69.5 [54 to 791.8] | 154.6 [123.8 to 247.1] | 202.5 [153.2 to 234.2]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  OC43-RBD-50 at Month 0-Total | 531.5 [300.8 to 1094.1] | 405 [238.8 to 827.1] | 502 [297.8 to 1111.4] | 664.5 [387.2 to 1143.9] | 534.1 [332.8 to 870.5]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  OC43-RBD-50 at Month 2-Total | 644.2 [240.1 to 1175.5] | 442.6 [256.7 to 1026.9] | 262.8 [209.5 to 2457] | 668 [491.3 to 975.8] | 708.8 [505.8 to 850.6]
  SARS-CoV-2 DB His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 DB His-250 at Month 0-Total | 309 [64.8 to 950.7] | 569 [185.1 to 1769.8] | 2676.2 [766.7 to 5780.2] | 1974.8 [654.8 to 4493] | 1454.8 [770.2 to 3669.6]
  SARS-CoV-2 DB His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 DB His-250 at Month 2-Total | 521.4 [254.1 to 1163.7] | 324.9 [119.4 to 602.3] | 1810.2 [706.5 to 2307.2] | 657.5 [140.2 to 1681.8] | 1577.5 [984 to 2064.1]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 DB His-50 at Month 0-Total | 1296.4 [279.2 to 3206.4] | 2033.8 [738.4 to 4901.8] | 8428.4 [2794.6 to 14028.2] | 5319.8 [1964 to 11542.6] | 5062.2 [2705.7 to 10498.8]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 DB His-50 at Month 2-Total | 2107.6 [1053.8 to 3960.2] | 1126.4 [479.2 to 2168.9] | 5008.8 [2829.2 to 6104.8] | 2415 [536.4 to 5368.4] | 3611.5 [3383.2 to 6262.4]
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 Nucleoprotein His-250 at Month 0-Total | 121.2 [67.4 to 398.9] | 348.6 [118.9 to 1087.1] | 1093.2 [619.8 to 2442.6] | 1485.8 [515.9 to 4719.9] | 569 [290.5 to 2004.9]
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 Nucleoprotein His-250 at Month 2-Total | 255.6 [138 to 602.1] | 163.1 [86.5 to 372.9] | 470.2 [161 to 1147.8] | 192.8 [118.4 to 743.3] | 352.5 [279.9 to 1082.9]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 542.1 [311.1 to 1765.8] | 1537 [531.3 to 4386.6] | 4777.8 [2256.8 to 9205.6] | 5562.5 [2107 to 13340.1] | 2238.2 [1168.5 to 7081]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 1070.2 [587.1 to 2268.8] | 654.1 [321.8 to 1547.6] | 1543 [641.8 to 3766.2] | 843.9 [444.6 to 2901.4] | 1432 [1016.4 to 3680.4]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 0-Total | 256.2 [16.3 to 1063.3] | 532.2 [181.1 to 1631.9] | 1957.4 [807.6 to 4744.6] | 1807.8 [470.1 to 4193.9] | 1579.6 [862.4 to 3270.7]
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S Hexapro_293F_PPF-250 at Month 2-Total | 875.8 [567.8 to 1584] | 254.2 [133.4 to 546.2] | 1378.5 [799.5 to 1757.5] | 495.2 [177.2 to 1190] | 961.2 [690.8 to 1517.4]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 1065.6 [78.1 to 3402.7] | 1990.8 [834.2 to 4490.6] | 4846 [2976.8 to 12278.4] | 5485 [1807.1 to 11671.9] | 5390.4 [3056.2 to 9709.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 3078.8 [2271.2 to 5186.6] | 1027.6 [604.2 to 1952.6] | 4093.8 [2869.2 to 5135.2] | 1839.9 [736.3 to 3652.6] | 3416.2 [2612.9 to 3548.5]
  SARS-CoV-2 S1 C His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1 C His-250 at Month 0-Total | 151.5 [28.1 to 669.1] | 408.2 [111.2 to 1447.3] | 1963.8 [513.2 to 4579.1] | 1399 [342.6 to 3522.9] | 1221.5 [513.7 to 3367.1]
  SARS-CoV-2 S1 C His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1 C His-250 at Month 2-Total | 323 [124.3 to 538.9] | 142.5 [48.1 to 319.6] | 924.2 [147 to 1186.2] | 392.6 [74.6 to 763.8] | 734.2 [547.9 to 1390.5]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 826.1 [99.6 to 2747.2] | 1619 [490 to 4896.8] | 6613.9 [2168 to 13021.4] | 4902.5 [1350.9 to 10810.8] | 4784.8 [2080.9 to 9906.1]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 1346.8 [525.9 to 2202.4] | 652.2 [224.8 to 1182.7] | 2569.5 [679.2 to 3422] | 1502.9 [287.5 to 3502.3] | 2455.5 [2061.9 to 4340.8]
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1S2 ECD His-250 at Month 0-Total | 352.6 [133.1 to 981.5] | 765.4 [330.4 to 1609.5] | 1606.1 [848.2 to 3024.8] | 1695.2 [862.9 to 3009.8] | 2312.9 [1082.8 to 4092.2]
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1S2 ECD His-250 at Month 2-Total | 991.2 [795.9 to 1138.3] | 885.5 [330.3 to 1514.1] | 1287.2 [1047 to 3310.8] | 989.9 [563.9 to 1424.7] | 1465.5 [1358 to 2566.9]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 1499.1 [552.9 to 3896.9] | 3341.1 [1419.6 to 6273.8] | 6263.9 [3477.1 to 10531.8] | 6482.2 [3425.2 to 10429.2] | 7607.4 [4498.7 to 12773]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 3985.6 [3313.5 to 4337.8] | 3409 [1285.3 to 4751.1] | 4357.2 [3539 to 9127.8] | 4217.1 [2144.5 to 5614.4] | 4748.8 [4172.8 to 7596.1]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 0-Total | 647 [59.8 to 1854.2] | 1215.1 [431.2 to 3214.7] | 4612.6 [1456.4 to 6742.9] | 3062.2 [1600.2 to 6567.4] | 3139 [1691.9 to 6339.6]
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 spike (PreS Nexelis)-250 at Month 2-Total | 2228.4 [1232 to 3540.6] | 622.6 [342.2 to 1149.2] | 2653.5 [1369.5 to 3131.2] | 1266.5 [555.8 to 2246.9] | 1792.5 [1722 to 3725]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 74 | 150 | 24 | 75 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 2660 [278.9 to 6524.4] | 4547.9 [1704.7 to 8595.2] | 10962.8 [5416.1 to 16444.4] | 9146.2 [4922.6 to 17148.5] | 10017.5 [6068.2 to 15630.2]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 7089.6 [4543.9 to 9975.9] | 2410 [1375.9 to 4038.2] | 6934.5 [4572.8 to 8524.5] | 3716.6 [2169.1 to 7332.9] | 5988.8 [5557.1 to 8848.6]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Total: number analyzed (Participants) | 64 | 91 | 15 | 62 | 43
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 0-Total | 51 [8.8 to 287.7] | 180.2 [41.6 to 551.8] | 1466.5 [411.2 to 4669.2] | 994.2 [322.2 to 2063.4] | 1004.5 [444.9 to 2333.9]
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2-NTD-AVI Biotin-250 at Month 2-Total | 46.2 [45.4 to 67.5] | 59.6 [22.4 to 158.1] | 353.8 [71.8 to 821.8] | 202.1 [92.1 to 347.4] | 774.2 [151.2 to 896.4]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 64 | 91 | 15 | 62 | 43
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 229.9 [46.7 to 1288.2] | 846.2 [192.2 to 2530.2] | 6049.8 [1836.8 to 12734.1] | 4312 [1477.6 to 8403.2] | 3966.5 [2065 to 9188.4]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 4 | 62 | 9 | 18 | 7
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 212.8 [202.1 to 299.2] | 255.6 [97.4 to 704.9] | 1390 [406.8 to 3060.2] | 825.1 [446.4 to 1427.5] | 2855.2 [646.1 to 3468.9]

22. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and COVID-19 Severity Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and COVID-19 severity
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  VRC7480_G614 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  VRC7480_G614 at Month 0-Peru | 25 | 56 | 17 | 41 | 28
  VRC7480_G614 at Month 0-Total: number analyzed (Participants) | 73 | 149 | 24 | 75 | 50
  VRC7480_G614 at Month 0-Total | 54 | 139 | 23 | 70 | 49
  VRC7480_G614 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 34 | 22
  VRC7480_G614 at Month 0-USA | 29 | 83 | 6 | 29 | 21
  VRC7480_G614 at Month 12-Peru: number analyzed (Participants) | 0 | 3 | 0 | 4 | 0
  VRC7480_G614 at Month 12-Peru |  | 3 |  | 4 |
  VRC7480_G614 at Month 12-Total: number analyzed (Participants) | 2 | 10 | 1 | 7 | 3
  VRC7480_G614 at Month 12-Total | 2 | 9 | 1 | 7 | 3
  VRC7480_G614 at Month 12-USA: number analyzed (Participants) | 2 | 7 | 1 | 3 | 3
  VRC7480_G614 at Month 12-USA | 2 | 6 | 1 | 3 | 3
  VRC7480_G614 at Month 2-Peru: number analyzed (Participants) | 19 | 36 | 15 | 30 | 6
  VRC7480_G614 at Month 2-Peru | 15 | 30 | 13 | 30 | 6
  VRC7480_G614 at Month 2-Total: number analyzed (Participants) | 36 | 98 | 18 | 47 | 17
  VRC7480_G614 at Month 2-Total | 29 | 84 | 16 | 45 | 17
  VRC7480_G614 at Month 2-USA: number analyzed (Participants) | 17 | 62 | 3 | 17 | 11
  VRC7480_G614 at Month 2-USA | 14 | 54 | 3 | 15 | 11
  VRC7480_G614 at Month 4-Peru: number analyzed (Participants) | 1 | 3 | 0 | 5 | 0
  VRC7480_G614 at Month 4-Peru | 1 | 3 |  | 5 |
  VRC7480_G614 at Month 4-Total: number analyzed (Participants) | 3 | 9 | 1 | 8 | 3
  VRC7480_G614 at Month 4-Total | 3 | 9 | 1 | 7 | 2
  VRC7480_G614 at Month 4-USA: number analyzed (Participants) | 2 | 6 | 1 | 3 | 3
  VRC7480_G614 at Month 4-USA | 2 | 6 | 1 | 2 | 2

23. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and COVID-19 Severity Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2,3,4, overall and by region and COVID-19 severity among America Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Titer
  VRC7480_G614-ID50 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  VRC7480_G614-ID50 at Month 0-Peru | 179.3 [68.2 to 544.4] | 527.7 [142.5 to 1636.1] | 2180 [635.6 to 4978] | 2826 [962.8 to 9093.1] | 2599 [750 to 5664.6]
  VRC7480_G614-ID50 at Month 0-Total: number analyzed (Participants) | 73 | 149 | 24 | 75 | 50
  VRC7480_G614-ID50 at Month 0-Total | 87.60 [5 to 340] | 284.8 [83.7 to 1078.9] | 1778 [702.2 to 4876.1] | 1497 [426.5 to 4781.4] | 1341 [524.2 to 4367.9]
  VRC7480_G614-ID50 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 34 | 22
  VRC7480_G614-ID50 at Month 0-USA | 53.00 [5 to 195] | 211.0 [66.1 to 627] | 1121 [875.7 to 3416.2] | 357.2 [190.8 to 1492.6] | 627.4 [373.5 to 1547.4]
  VRC7480_G614-ID50 at Month 12-Peru: number analyzed (Participants) | 0 | 3 | 0 | 4 | 0
  VRC7480_G614-ID50 at Month 12-Peru |  | 289.6 [177.4 to 578.1] |  | 305.6 [97.2 to 609.4] |
  VRC7480_G614-ID50 at Month 12-Total: number analyzed (Participants) | 2 | 10 | 1 | 7 | 3
  VRC7480_G614-ID50 at Month 12-Total | 220.4 [157.3 to 283.4] | 285.7 [61.5 to 682.6] | 726.3 [726.3 to 726.3] | 411.9 [119 to 460.7] | 232.2 [172.7 to 239]
  VRC7480_G614-ID50 at Month 12-USA: number analyzed (Participants) | 2 | 7 | 1 | 3 | 3
  VRC7480_G614-ID50 at Month 12-USA | 220.4 [157.3 to 283.4] | 281.8 [59.6 to 658] | 726.3 [726.3 to 726.3] | 411.9 [264.9 to 421.2] | 232.2 [172.7 to 239]
  VRC7480_G614-ID50 at Month 2-Peru: number analyzed (Participants) | 19 | 36 | 15 | 30 | 6
  VRC7480_G614-ID50 at Month 2-Peru | 35.10 [10 to 56.2] | 81.00 [10 to 189.2] | 335.2 [74.7 to 643.1] | 663.0 [281.9 to 1059.3] | 281.9 [222.4 to 367.7]
  VRC7480_G614-ID50 at Month 2-Total: number analyzed (Participants) | 36 | 98 | 18 | 47 | 17
  VRC7480_G614-ID50 at Month 2-Total | 38.30 [10 to 82] | 85.40 [35.8 to 202.9] | 338.8 [65 to 832.1] | 358.0 [205.1 to 843.3] | 325.7 [165.2 to 564.2]
  VRC7480_G614-ID50 at Month 2-USA: number analyzed (Participants) | 17 | 62 | 3 | 17 | 11
  VRC7480_G614-ID50 at Month 2-USA | 47.30 [25.1 to 106.7] | 89.90 [37.5 to 214.7] | 890.3 [471.8 to 1046.2] | 176.8 [28.6 to 358] | 436.3 [121.5 to 872.7]
  VRC7480_G614-ID50 at Month 4-Peru: number analyzed (Participants) | 1 | 3 | 0 | 5 | 0
  VRC7480_G614-ID50 at Month 4-Peru | 113.2 [113.2 to 113.2] | 60.30 [44.8 to 146.2] |  | 245.7 [151.7 to 411.9] |
  VRC7480_G614-ID50 at Month 4-Total: number analyzed (Participants) | 3 | 9 | 1 | 8 | 3
  VRC7480_G614-ID50 at Month 4-Total | 253.3 [183.2 to 489.8] | 117.8 [60.3 to 232.2] | 1034.5 [1034.5 to 1034.5] | 198.7 [111.4 to 461.1] | 281.8 [143.4 to 314.1]
  VRC7480_G614-ID50 at Month 4-USA: number analyzed (Participants) | 2 | 6 | 1 | 3 | 3
  VRC7480_G614-ID50 at Month 4-USA | 489.8 [371.5 to 608] | 152.4 [100.2 to 382.5] | 1034.5 [1034.5 to 1034.5] | 120.2 [62.6 to 419.6] | 281.8 [143.4 to 314.1]
  VRC7480_G614-ID80 at Month 0-Peru: number analyzed (Participants) | 29 | 61 | 18 | 41 | 28
  VRC7480_G614-ID80 at Month 0-Peru | 42.50 [25.5 to 132.4] | 117.6 [39.2 to 354.1] | 459.3 [159.2 to 799.7] | 601.8 [244.5 to 1101.3] | 675.6 [205 to 1113]
  VRC7480_G614-ID80 at Month 0-Total: number analyzed (Participants) | 73 | 149 | 24 | 75 | 50
  VRC7480_G614-ID80 at Month 0-Total | 27.90 [5 to 70] | 60.10 [27.5 to 209] | 321.5 [161.2 to 729.1] | 262.4 [135.6 to 821.4] | 293.9 [136.2 to 890.6]
  VRC7480_G614-ID80 at Month 0-USA: number analyzed (Participants) | 44 | 88 | 6 | 34 | 22
  VRC7480_G614-ID80 at Month 0-USA | 20.20 [5 to 51.2] | 41.40 [21.6 to 144.8] | 227.0 [185.8 to 537.5] | 127.3 [62.6 to 266.1] | 169.2 [108 to 343.9]
  VRC7480_G614-ID80 at Month 12-Peru: number analyzed (Participants) | 0 | 3 | 0 | 4 | 0
  VRC7480_G614-ID80 at Month 12-Peru |  | 104.3 [75.2 to 181.7] |  | 91.00 [36.8 to 198.4] |
  VRC7480_G614-ID80 at Month 12-Total: number analyzed (Participants) | 2 | 10 | 1 | 7 | 3
  VRC7480_G614-ID80 at Month 12-Total | 75.50 [53.1 to 98] | 107.9 [29.8 to 187.6] | 185.8 [185.8 to 185.8] | 128.3 [45.4 to 146.9] | 73.50 [55.4 to 80.4]
  VRC7480_G614-ID80 at Month 12-USA: number analyzed (Participants) | 2 | 7 | 1 | 3 | 3
  VRC7480_G614-ID80 at Month 12-USA | 75.50 [53.1 to 98] | 111.5 [15.9 to 185.8] | 185.8 [185.8 to 185.8] | 128.3 [86.2 to 143.4] | 73.50 [55.4 to 80.4]
  VRC7480_G614-ID80 at Month 2-Peru: number analyzed (Participants) | 19 | 36 | 15 | 30 | 6
  VRC7480_G614-ID80 at Month 2-Peru | 10.00 [10 to 25.1] | 28.50 [10 to 56.1] | 103.4 [27.1 to 173] | 190.3 [113.3 to 310.5] | 124.3 [73 to 141.1]
  VRC7480_G614-ID80 at Month 2-Total: number analyzed (Participants) | 36 | 98 | 18 | 47 | 17
  VRC7480_G614-ID80 at Month 2-Total | 10.00 [10 to 31.4] | 28.50 [10 to 57.2] | 109.7 [26.4 to 232.8] | 127.8 [62 to 237.9] | 120.6 [55.7 to 172.8]
  VRC7480_G614-ID80 at Month 2-USA: number analyzed (Participants) | 17 | 62 | 3 | 17 | 11
  VRC7480_G614-ID80 at Month 2-USA | 13.70 [10 to 38.4] | 29.00 [10 to 56.4] | 246.1 [134.1 to 296.1] | 54.10 [10 to 82.1] | 120.4 [45.1 to 223.5]
  VRC7480_G614-ID80 at Month 4-Peru: number analyzed (Participants) | 1 | 3 | 0 | 5 | 0
  VRC7480_G614-ID80 at Month 4-Peru | 37.30 [37.3 to 37.3] | 13.70 [10.6 to 50.5] |  | 73.50 [55.7 to 158.5] |
  VRC7480_G614-ID80 at Month 4-Total: number analyzed (Participants) | 3 | 9 | 1 | 8 | 3
  VRC7480_G614-ID80 at Month 4-Total | 80.70 [59 to 133.2] | 44.10 [24.4 to 87.3] | 334.0 [334 to 334] | 64.60 [42.6 to 163.1] | 111.5 [58.3 to 116]
  VRC7480_G614-ID80 at Month 4-USA: number analyzed (Participants) | 2 | 6 | 1 | 3 | 3
  VRC7480_G614-ID80 at Month 4-USA | 133.2 [107 to 159.5] | 53.40 [34 to 111.5] | 334.0 [334 to 334] | 46.60 [25.8 to 111.8] | 111.5 [58.3 to 116]

24. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and COVID-19 Severity Among Africa Cohort
Description: as for outcome 22
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Group 6: Hospitalized, ICU and ECMO
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 96 | 161 | 26 | 67 | 21 | 1
Participants
  SARS-Cov-2 D614G at Month 0-RSA: number analyzed (Participants) | 65 | 114 | 21 | 30 | 8 | 1
  SARS-Cov-2 D614G at Month 0-RSA | 59 | 107 | 19 | 28 | 8 | 1
  SARS-Cov-2 D614G at Month 0-Total: number analyzed (Participants) | 83 | 152 | 25 | 47 | 15 | 1
  SARS-Cov-2 D614G at Month 0-Total | 73 | 137 | 22 | 44 | 15 | 1
  SARS-Cov-2 D614G at Month 0-non-RSA: number analyzed (Participants) | 18 | 38 | 4 | 17 | 7 | 0
  SARS-Cov-2 D614G at Month 0-non-RSA | 14 | 30 | 3 | 16 | 7 |
  SARS-Cov-2 D614G at Month 12-RSA: number analyzed (Participants) | 34 | 47 | 12 | 14 | 5 | 0
  SARS-Cov-2 D614G at Month 12-RSA | 33 | 46 | 12 | 14 | 5 |
  SARS-Cov-2 D614G at Month 12-Total: number analyzed (Participants) | 51 | 80 | 14 | 28 | 8 | 0
  SARS-Cov-2 D614G at Month 12-Total | 49 | 78 | 14 | 27 | 8 |
  SARS-Cov-2 D614G at Month 12-non-RSA: number analyzed (Participants) | 17 | 33 | 2 | 14 | 3 | 0
  SARS-Cov-2 D614G at Month 12-non-RSA | 16 | 32 | 2 | 13 | 3 |
  SARS-Cov-2 D614G at Month 2-RSA: number analyzed (Participants) | 40 | 77 | 16 | 18 | 6 | 1
  SARS-Cov-2 D614G at Month 2-RSA | 36 | 72 | 15 | 18 | 6 | 1
  SARS-Cov-2 D614G at Month 2-Total: number analyzed (Participants) | 58 | 112 | 20 | 36 | 10 | 1
  SARS-Cov-2 D614G at Month 2-Total | 50 | 97 | 19 | 35 | 10 | 1
  SARS-Cov-2 D614G at Month 2-non-RSA: number analyzed (Participants) | 18 | 35 | 4 | 18 | 4 | 0
  SARS-Cov-2 D614G at Month 2-non-RSA | 14 | 25 | 4 | 17 | 4 |
  SARS-Cov-2 D614G at Month 4-RSA: number analyzed (Participants) | 41 | 77 | 16 | 17 | 5 | 1
  SARS-Cov-2 D614G at Month 4-RSA | 37 | 70 | 15 | 16 | 5 | 1
  SARS-Cov-2 D614G at Month 4-Total: number analyzed (Participants) | 57 | 107 | 19 | 34 | 10 | 1
  SARS-Cov-2 D614G at Month 4-Total | 52 | 96 | 18 | 31 | 10 | 1
  SARS-Cov-2 D614G at Month 4-non-RSA: number analyzed (Participants) | 16 | 30 | 3 | 17 | 5 | 0
  SARS-Cov-2 D614G at Month 4-non-RSA | 15 | 26 | 3 | 15 | 5 |

25. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and COVID-19 Severity Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and COVID-19 severity among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 96 | 161 | 26 | 67 | 21 | 1
Titer
  SARS-Cov-2 D614G-ID50 at Month 0-RSA: number analyzed (Participants) | 65 | 114 | 21 | 30 | 8 | 1
  SARS-Cov-2 D614G-ID50 at Month 0-RSA | 189.0 [49.2 to 474.5] | 344.8 [132.7 to 1342.9] | 422.3 [172.5 to 932.1] | 1136 [283.4 to 2206.3] | 1594 [464.4 to 3441.6] | 2658.5 [2658.5 to 2658.5]
  SARS-Cov-2 D614G-ID50 at Month 0-Total: number analyzed (Participants) | 83 | 152 | 25 | 47 | 15 | 1
  SARS-Cov-2 D614G-ID50 at Month 0-Total | 183.5 [40.7 to 361.5] | 327.3 [101.2 to 1157.5] | 397.0 [112.5 to 851.1] | 1304 [227.8 to 2076.4] | 1672 [575.1 to 3064] | 2658.5 [2658.5 to 2658.5]
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA: number analyzed (Participants) | 18 | 38 | 4 | 17 | 7 | 0
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA | 74.20 [8.2 to 216.8] | 265.1 [19.3 to 714.1] | 80.60 [37.7 to 243.9] | 1328 [144.8 to 1786.8] | 1672 [1086.5 to 2746.1] |
  SARS-Cov-2 D614G-ID50 at Month 12-RSA: number analyzed (Participants) | 34 | 47 | 12 | 14 | 5 | 0
  SARS-Cov-2 D614G-ID50 at Month 12-RSA | 374.2 [120.2 to 3956.1] | 2543 [425.3 to 9673.3] | 1558 [361.6 to 4887.3] | 12337 [4219 to 37945.2] | 2700 [1430.6 to 5603.8] |
  SARS-Cov-2 D614G-ID50 at Month 12-Total: number analyzed (Participants) | 51 | 80 | 14 | 28 | 8 | 0
  SARS-Cov-2 D614G-ID50 at Month 12-Total | 559.2 [177.1 to 2693.7] | 997.3 [291.7 to 7868.9] | 1558 [442 to 5741.1] | 5130 [430.3 to 19363] | 2065 [1131.6 to 6481.4] |
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA: number analyzed (Participants) | 17 | 33 | 2 | 14 | 3 | 0
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA | 1160 [337 to 2281.9] | 478.9 [239.6 to 3393.2] | 3521 [2196.6 to 4845.7] | 1522 [306.6 to 6278.1] | 265.6 [237.3 to 4690] |
  SARS-Cov-2 D614G-ID50 at Month 2-RSA: number analyzed (Participants) | 40 | 77 | 16 | 18 | 6 | 1
  SARS-Cov-2 D614G-ID50 at Month 2-RSA | 86.30 [10 to 231.2] | 165.4 [59.9 to 586.1] | 224.8 [76.7 to 535.8] | 540.6 [185.2 to 1287.9] | 827.2 [337.9 to 1283.4] | 1925.3 [1925.3 to 1925.3]
  SARS-Cov-2 D614G-ID50 at Month 2-Total: number analyzed (Participants) | 58 | 112 | 20 | 36 | 10 | 1
  SARS-Cov-2 D614G-ID50 at Month 2-Total | 68.40 [10 to 198] | 125.3 [43.5 to 413.3] | 211.4 [67.7 to 451.1] | 490.0 [110.6 to 963.2] | 494.6 [115.5 to 884.7] | 1925.3 [1925.3 to 1925.3]
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA: number analyzed (Participants) | 18 | 35 | 4 | 18 | 4 | 0
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA | 51.90 [8.7 to 139.6] | 52.40 [5 to 192.2] | 130.2 [48.1 to 211.4] | 427.5 [50.8 to 834.3] | 157.3 [80.1 to 385.8] |
  SARS-Cov-2 D614G-ID50 at Month 4-RSA: number analyzed (Participants) | 41 | 77 | 16 | 17 | 5 | 1
  SARS-Cov-2 D614G-ID50 at Month 4-RSA | 203.6 [48.5 to 552.1] | 356.5 [83.7 to 932.5] | 382.2 [101.8 to 619.6] | 657.1 [214.5 to 1422.1] | 738.7 [239.1 to 1161.9] | 2231.7 [2231.7 to 2231.7]
  SARS-Cov-2 D614G-ID50 at Month 4-Total: number analyzed (Participants) | 57 | 107 | 19 | 34 | 10 | 1
  SARS-Cov-2 D614G-ID50 at Month 4-Total | 148.5 [54.3 to 314.9] | 276.5 [71.8 to 880.5] | 251.2 [93.2 to 531.6] | 713.2 [220.9 to 1403.5] | 659.8 [267.7 to 1110] | 2231.7 [2231.7 to 2231.7]
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA: number analyzed (Participants) | 16 | 30 | 3 | 17 | 5 | 0
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA | 130.8 [71.1 to 168.6] | 174.1 [42.5 to 392.4] | 95.10 [83.3 to 165] | 1114 [333.2 to 1310.4] | 580.8 [353.6 to 954.2] |
  SARS-Cov-2 D614G-ID80 at Month 0-RSA: number analyzed (Participants) | 65 | 114 | 21 | 30 | 8 | 1
  SARS-Cov-2 D614G-ID80 at Month 0-RSA | 42.50 [10 to 130.6] | 88.50 [35.1 to 314.8] | 100.9 [37.3 to 238.5] | 303.0 [83.1 to 573.9] | 328.1 [129.5 to 571.4] | 813.8 [813.8 to 813.8]
  SARS-Cov-2 D614G-ID80 at Month 0-Total: number analyzed (Participants) | 83 | 152 | 25 | 47 | 15 | 1
  SARS-Cov-2 D614G-ID80 at Month 0-Total | 40.40 [10 to 111.3] | 80.40 [31.7 to 240.8] | 83.20 [30.9 to 202.6] | 347.3 [65.3 to 605.8] | 399.5 [149.6 to 715.7] | 813.8 [813.8 to 813.8]
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA: number analyzed (Participants) | 18 | 38 | 4 | 17 | 7 | 0
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA | 27.10 [7.5 to 46.6] | 45.70 [10 to 181.3] | 27.50 [19.1 to 65.1] | 361.0 [43.1 to 615.2] | 614.9 [247.2 to 836.2] |
  SARS-Cov-2 D614G-ID80 at Month 12-RSA: number analyzed (Participants) | 34 | 47 | 12 | 14 | 5 | 0
  SARS-Cov-2 D614G-ID80 at Month 12-RSA | 122.4 [36 to 894.2] | 634.9 [116.7 to 2755] | 391.2 [126.8 to 1189.4] | 3390 [1041.9 to 5450.3] | 452.5 [389.6 to 1378.9] |
  SARS-Cov-2 D614G-ID80 at Month 12-Total: number analyzed (Participants) | 51 | 80 | 14 | 28 | 8 | 0
  SARS-Cov-2 D614G-ID80 at Month 12-Total | 161.2 [41.9 to 776.1] | 240.7 [104.8 to 2149.5] | 391.2 [154.3 to 1287.7] | 1914 [170 to 4128.4] | 421.0 [242 to 1681.1] |
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA: number analyzed (Participants) | 17 | 33 | 2 | 14 | 3 | 0
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA | 381.6 [92.4 to 712.6] | 161.8 [70.6 to 793.1] | 797.9 [518.3 to 1077.5] | 413.3 [131.4 to 2113.3] | 100.0 [81.4 to 1343.8] |
  SARS-Cov-2 D614G-ID80 at Month 2-RSA: number analyzed (Participants) | 40 | 77 | 16 | 18 | 6 | 1
  SARS-Cov-2 D614G-ID80 at Month 2-RSA | 31.70 [10 to 47.1] | 43.10 [20.7 to 173.5] | 65.00 [31 to 166.6] | 142.4 [63.7 to 230.7] | 203.1 [97.5 to 320.8] | 678.1 [678.1 to 678.1]
  SARS-Cov-2 D614G-ID80 at Month 2-Total: number analyzed (Participants) | 58 | 112 | 20 | 36 | 10 | 1
  SARS-Cov-2 D614G-ID80 at Month 2-Total | 22.70 [10 to 40.9] | 36.10 [10 to 122] | 53.00 [29.6 to 118.7] | 137.1 [37 to 207.6] | 146.1 [36.7 to 204.8] | 678.1 [678.1 to 678.1]
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA: number analyzed (Participants) | 18 | 35 | 4 | 18 | 4 | 0
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA | 10.00 [7.5 to 24.3] | 22.30 [5 to 42.7] | 31.50 [10 to 53] | 114.1 [16.3 to 196.7] | 65.20 [27.1 to 124.4] |
  SARS-Cov-2 D614G-ID80 at Month 4-RSA: number analyzed (Participants) | 41 | 77 | 16 | 17 | 5 | 1
  SARS-Cov-2 D614G-ID80 at Month 4-RSA | 42.30 [10 to 152.9] | 102.1 [28.8 to 226] | 101.1 [33.8 to 167.5] | 169.7 [63.4 to 562.3] | 209.9 [60.9 to 274.8] | 643.1 [643.1 to 643.1]
  SARS-Cov-2 D614G-ID80 at Month 4-Total: number analyzed (Participants) | 57 | 107 | 19 | 34 | 10 | 1
  SARS-Cov-2 D614G-ID80 at Month 4-Total | 36.50 [10 to 120.5] | 85.60 [24.1 to 202.1] | 64.80 [33 to 152.5] | 179.1 [70.7 to 552.4] | 193.5 [65.9 to 264.7] | 643.1 [643.1 to 643.1]
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA: number analyzed (Participants) | 16 | 30 | 3 | 17 | 5 | 0
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA | 34.00 [22.4 to 41] | 46.10 [13.5 to 140.2] | 32.50 [30.7 to 43.9] | 239.3 [118 to 353.5] | 177.1 [80.8 to 234.7] |

26. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (ADCC) by Region and COVID-19 Severity Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by antibody-dependent cellular cytotoxicity assay (ADCC) at Visit 1, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru: number analyzed (Participants) | 24 | 47 | 12 | 34 | 11
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru | 10 | 32 | 8 | 31 | 11
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 58 | 99 | 16 | 57 | 26
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 15 | 53 | 11 | 49 | 24
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA: number analyzed (Participants) | 34 | 52 | 4 | 23 | 15
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA | 5 | 21 | 3 | 18 | 13
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru: number analyzed (Participants) | 24 | 47 | 12 | 34 | 11
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru | 10 | 34 | 10 | 31 | 10
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 58 | 99 | 16 | 57 | 26
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 17 | 59 | 13 | 46 | 18
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA: number analyzed (Participants) | 34 | 52 | 4 | 23 | 15
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA | 7 | 25 | 3 | 15 | 8

27. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (ADCC) by Region and COVID-19 Severity Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by antibody-dependent cellular cytotoxicity assay (ADCC) Visit 1, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: Percent CD107a+ NK Cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Percent CD107a+ NK Cells
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru: number analyzed (Participants) | 24 | 47 | 12 | 34 | 11
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Peru | 1.6 [0.5 to 4.6] | 7.7 [3.3 to 13.8] | 11.3 [2.8 to 21.1] | 13.6 [9.5 to 15.7] | 17.9 [11.7 to 26]
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 58 | 99 | 16 | 57 | 26
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 1.1 [0 to 4] | 4.6 [1.4 to 9] | 10.8 [3.8 to 17.1] | 13.3 [6.6 to 15.9] | 17.6 [11.6 to 22]
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA: number analyzed (Participants) | 34 | 52 | 4 | 23 | 15
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-USA | 0.7 [0 to 2.3] | 3.4 [1.1 to 6.7] | 9.5 [5.9 to 13.3] | 10.8 [5.6 to 16.6] | 17.5 [11.7 to 20.3]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru: number analyzed (Participants) | 24 | 47 | 12 | 34 | 11
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Peru | 4.8 [2.2 to 11] | 8.6 [4.1 to 12.3] | 12.9 [8.3 to 15] | 15.9 [12.3 to 18.3] | 11.8 [9.2 to 16.8]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 58 | 99 | 16 | 57 | 26
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 3.8 [0.2 to 6] | 6 [3.5 to 11.2] | 12 [6.6 to 13.8] | 13.1 [7.6 to 16.7] | 9.5 [3.5 to 14.1]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA: number analyzed (Participants) | 34 | 52 | 4 | 23 | 15
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-USA | 1.6 [0 to 5.1] | 5.2 [3 to 7.5] | 7 [5.1 to 9.5] | 9.4 [3 to 12.7] | 5.9 [2.2 to 12.2]

28. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate (ICS) by Region and COVID-19 Severity Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate by flow cytometry at Visit 1, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
Participants
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD4+-Any COV2 at Month 0-Peru | 15 | 46 | 14 | 40 | 28
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 71 | 147 | 23 | 75 | 49
  CD4+-Any COV2 at Month 0-Total | 33 | 107 | 19 | 67 | 46
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 43 | 85 | 6 | 34 | 21
  CD4+-Any COV2 at Month 0-USA | 18 | 61 | 5 | 27 | 18
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 27 | 62 | 17 | 40 | 28
  CD4+-E M at Month 0-Peru | 7 | 35 | 12 | 34 | 27
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 68 | 146 | 22 | 73 | 49
  CD4+-E M at Month 0-Total | 16 | 72 | 14 | 58 | 43
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 41 | 84 | 5 | 33 | 21
  CD4+-E M at Month 0-USA | 9 | 37 | 2 | 24 | 16
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD4+-N at Month 0-Peru | 11 | 37 | 12 | 31 | 25
  CD4+-N at Month 0-Total: number analyzed (Participants) | 70 | 147 | 23 | 75 | 49
  CD4+-N at Month 0-Total | 20 | 87 | 16 | 56 | 42
  CD4+-N at Month 0-USA: number analyzed (Participants) | 42 | 85 | 6 | 34 | 21
  CD4+-N at Month 0-USA | 9 | 50 | 4 | 25 | 17
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 28 | 61 | 17 | 39 | 27
  CD4+-ORF3a6 at Month 0-Peru | 3 | 22 | 5 | 20 | 15
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 69 | 146 | 22 | 72 | 48
  CD4+-ORF3a6 at Month 0-Total | 8 | 42 | 8 | 42 | 26
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 41 | 85 | 5 | 33 | 21
  CD4+-ORF3a6 at Month 0-USA | 5 | 20 | 3 | 22 | 11
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 40 | 27
  CD4+-ORF7a7b8 at Month 0-Peru | 5 | 23 | 7 | 30 | 21
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 68 | 145 | 23 | 72 | 48
  CD4+-ORF7a7b8 at Month 0-Total | 9 | 45 | 10 | 46 | 32
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 40 | 83 | 6 | 32 | 21
  CD4+-ORF7a7b8 at Month 0-USA | 4 | 22 | 3 | 16 | 11
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 27 | 61 | 17 | 40 | 28
  CD4+-S1 at Month 0-Peru | 10 | 37 | 14 | 38 | 27
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 70 | 146 | 23 | 74 | 48
  CD4+-S1 at Month 0-Total | 20 | 84 | 19 | 64 | 44
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 43 | 85 | 6 | 34 | 20
  CD4+-S1 at Month 0-USA | 10 | 47 | 5 | 26 | 17
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD4+-S2 at Month 0-Peru | 12 | 32 | 11 | 34 | 27
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 71 | 147 | 23 | 75 | 49
  CD4+-S2 at Month 0-Total | 21 | 78 | 16 | 59 | 45
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 43 | 85 | 6 | 34 | 21
  CD4+-S2 at Month 0-USA | 9 | 46 | 5 | 25 | 18
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD4+-Spike at Month 0-Peru | 13 | 40 | 14 | 40 | 28
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 71 | 147 | 23 | 75 | 49
  CD4+-Spike at Month 0-Total | 25 | 96 | 19 | 66 | 46
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 43 | 85 | 6 | 34 | 21
  CD4+-Spike at Month 0-USA | 12 | 56 | 5 | 26 | 18
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD8+-Any COV2 at Month 0-Peru | 14 | 41 | 10 | 34 | 23
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 71 | 146 | 23 | 75 | 49
  CD8+-Any COV2 at Month 0-Total | 33 | 93 | 16 | 54 | 36
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 43 | 84 | 6 | 34 | 21
  CD8+-Any COV2 at Month 0-USA | 19 | 52 | 6 | 20 | 13
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 40 | 28
  CD8+-E M at Month 0-Peru | 0 | 1 | 0 | 7 | 5
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 69 | 145 | 22 | 73 | 49
  CD8+-E M at Month 0-Total | 3 | 8 | 2 | 10 | 7
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 41 | 83 | 5 | 33 | 21
  CD8+-E M at Month 0-USA | 3 | 7 | 2 | 3 | 2
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD8+-N at Month 0-Peru | 11 | 39 | 8 | 30 | 20
  CD8+-N at Month 0-Total: number analyzed (Participants) | 70 | 146 | 23 | 75 | 49
  CD8+-N at Month 0-Total | 27 | 84 | 13 | 46 | 30
  CD8+-N at Month 0-USA: number analyzed (Participants) | 42 | 84 | 6 | 34 | 21
  CD8+-N at Month 0-USA | 16 | 45 | 5 | 16 | 10
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 40 | 27
  CD8+-ORF3a6 at Month 0-Peru | 4 | 16 | 3 | 18 | 9
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 69 | 146 | 22 | 73 | 48
  CD8+-ORF3a6 at Month 0-Total | 8 | 29 | 6 | 25 | 12
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 41 | 84 | 5 | 33 | 21
  CD8+-ORF3a6 at Month 0-USA | 4 | 13 | 3 | 7 | 3
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 40 | 27
  CD8+-ORF7a7b8 at Month 0-Peru | 3 | 17 | 3 | 17 | 11
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 67 | 144 | 23 | 72 | 48
  CD8+-ORF7a7b8 at Month 0-Total | 6 | 23 | 5 | 22 | 15
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 39 | 82 | 6 | 32 | 21
  CD8+-ORF7a7b8 at Month 0-USA | 3 | 6 | 2 | 5 | 4
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 27 | 62 | 17 | 40 | 28
  CD8+-S1 at Month 0-Peru | 1 | 14 | 5 | 12 | 10
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 70 | 146 | 23 | 74 | 48
  CD8+-S1 at Month 0-Total | 1 | 33 | 8 | 15 | 14
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 43 | 84 | 6 | 34 | 20
  CD8+-S1 at Month 0-USA | 0 | 19 | 3 | 3 | 4
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 40 | 28
  CD8+-S2 at Month 0-Peru | 3 | 4 | 2 | 4 | 5
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 71 | 146 | 23 | 74 | 49
  CD8+-S2 at Month 0-Total | 4 | 11 | 3 | 5 | 7
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 43 | 84 | 6 | 34 | 21
  CD8+-S2 at Month 0-USA | 1 | 7 | 1 | 1 | 2
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 28 | 62 | 17 | 41 | 28
  CD8+-Spike at Month 0-Peru | 4 | 15 | 5 | 12 | 11
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 71 | 146 | 23 | 75 | 49
  CD8+-Spike at Month 0-Total | 5 | 38 | 8 | 15 | 16
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 43 | 84 | 6 | 34 | 21
  CD8+-Spike at Month 0-USA | 1 | 23 | 3 | 3 | 5

29. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude (ICS) by Region and COVID-19 Severity Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and COVID-19 severity among America Cohort
Time Frame: Measured at Months 0
Population: American Population with positive responders (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: % T cells expressing IFN-g/IL-2
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
% T cells expressing IFN-g/IL-2
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 15 | 46 | 14 | 40 | 28
  CD4+-Any COV2 at Month 0-Peru | 0.2 [0.2 to 0.4] | 0.6 [0.3 to 1.2] | 0.5 [0.4 to 0.7] | 1.1 [0.6 to 1.6] | 1.1 [0.6 to 1.8]
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 33 | 107 | 19 | 67 | 46
  CD4+-Any COV2 at Month 0-Total | 0.3 [0.2 to 0.5] | 0.4 [0.3 to 0.9] | 0.5 [0.4 to 0.7] | 1 [0.6 to 1.4] | 1 [0.6 to 1.4]
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 18 | 61 | 5 | 27 | 18
  CD4+-Any COV2 at Month 0-USA | 0.3 [0.1 to 0.6] | 0.4 [0.3 to 0.6] | 0.7 [0.6 to 1.8] | 0.8 [0.5 to 1.1] | 0.9 [0.6 to 1.1]
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 7 | 35 | 12 | 34 | 27
  CD4+-E M at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.1] | 0.3 [0.2 to 0.4] | 0.2 [0.2 to 0.4]
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 16 | 72 | 14 | 58 | 43
  CD4+-E M at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 9 | 37 | 2 | 24 | 16
  CD4+-E M at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 11 | 37 | 12 | 31 | 25
  CD4+-N at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD4+-N at Month 0-Total: number analyzed (Participants) | 20 | 87 | 16 | 56 | 42
  CD4+-N at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-USA: number analyzed (Participants) | 9 | 50 | 4 | 25 | 17
  CD4+-N at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.3 [0.1 to 0.7] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 3 | 22 | 5 | 20 | 15
  CD4+-ORF3a6 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 8 | 42 | 8 | 42 | 26
  CD4+-ORF3a6 at Month 0-Total | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 5 | 20 | 3 | 22 | 11
  CD4+-ORF3a6 at Month 0-USA | 0.3 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 5 | 23 | 7 | 30 | 21
  CD4+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 9 | 45 | 10 | 46 | 32
  CD4+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 4 | 22 | 3 | 16 | 11
  CD4+-ORF7a7b8 at Month 0-USA | 0.1 [0 to 0.1] | 0.1 [0 to 0.1] | 0.2 [0.2 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 10 | 37 | 14 | 38 | 27
  CD4+-S1 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.4 [0.2 to 0.5] | 0.4 [0.2 to 0.6]
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 20 | 84 | 19 | 64 | 44
  CD4+-S1 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.4] | 0.3 [0.2 to 0.4]
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 10 | 47 | 5 | 26 | 17
  CD4+-S1 at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.7] | 0.2 [0.2 to 0.3] | 0.3 [0.2 to 0.3]
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 12 | 32 | 11 | 34 | 27
  CD4+-S2 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.4]
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 21 | 78 | 16 | 59 | 45
  CD4+-S2 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 9 | 46 | 5 | 25 | 18
  CD4+-S2 at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.2]
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 13 | 40 | 14 | 40 | 28
  CD4+-Spike at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.3] | 0.5 [0.2 to 0.7] | 0.6 [0.3 to 0.8]
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 25 | 96 | 19 | 66 | 46
  CD4+-Spike at Month 0-Total | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.4 [0.2 to 0.6] | 0.5 [0.3 to 0.7]
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 12 | 56 | 5 | 26 | 18
  CD4+-Spike at Month 0-USA | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.9] | 0.3 [0.2 to 0.6] | 0.4 [0.3 to 0.5]
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 14 | 41 | 10 | 34 | 23
  CD8+-Any COV2 at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.5 [0.3 to 1] | 0.4 [0.2 to 0.5] | 0.9 [0.3 to 2.2] | 0.6 [0.3 to 1.2]
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 33 | 93 | 16 | 54 | 36
  CD8+-Any COV2 at Month 0-Total | 0.2 [0.1 to 0.3] | 0.4 [0.2 to 0.7] | 0.4 [0.2 to 1] | 0.6 [0.2 to 1.6] | 0.5 [0.3 to 1.1]
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 19 | 52 | 6 | 20 | 13
  CD8+-Any COV2 at Month 0-USA | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.7] | 0.6 [0.3 to 1.5] | 0.3 [0.1 to 0.6] | 0.5 [0.3 to 0.8]
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 7 | 5
  CD8+-E M at Month 0-Peru |  | 0.1 [0.1 to 0.1] |  | 0.2 [0.2 to 0.2] | 0.2 [0.1 to 0.2]
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 3 | 8 | 2 | 10 | 7
  CD8+-E M at Month 0-Total | 0.2 [0.1 to 1.2] | 0.1 [0.1 to 0.2] | 0.4 [0.2 to 0.5] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 3 | 7 | 2 | 3 | 2
  CD8+-E M at Month 0-USA | 0.2 [0.1 to 1.2] | 0.1 [0.1 to 0.2] | 0.4 [0.2 to 0.5] | 0.1 [0.1 to 0.1] | 0.4 [0.3 to 0.6]
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 11 | 39 | 8 | 30 | 20
  CD8+-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.3 [0.1 to 0.5] | 0.2 [0.1 to 0.3] | 0.5 [0.2 to 1.2] | 0.2 [0.1 to 0.9]
  CD8+-N at Month 0-Total: number analyzed (Participants) | 27 | 84 | 13 | 46 | 30
  CD8+-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 1.1] | 0.2 [0.2 to 0.8]
  CD8+-N at Month 0-USA: number analyzed (Participants) | 16 | 45 | 5 | 16 | 10
  CD8+-N at Month 0-USA | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.6 [0.3 to 0.6] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.6]
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 4 | 16 | 3 | 18 | 9
  CD8+-ORF3a6 at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.4 [0.2 to 0.4] | 0.4 [0.1 to 0.8] | 0.2 [0.1 to 0.6]
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 8 | 29 | 6 | 25 | 12
  CD8+-ORF3a6 at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.6] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 4 | 13 | 3 | 7 | 3
  CD8+-ORF3a6 at Month 0-USA | 0.1 [0.1 to 0.2] | 0.3 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.2 to 0.2]
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 3 | 17 | 3 | 17 | 11
  CD8+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.4 [0.2 to 0.5] | 0.7 [0.2 to 0.9] | 0.2 [0.1 to 0.6]
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 6 | 23 | 5 | 22 | 15
  CD8+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.6 [0.2 to 0.8] | 0.2 [0.1 to 0.4]
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 3 | 6 | 2 | 5 | 4
  CD8+-ORF7a7b8 at Month 0-USA | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.1] | 0.5 [0.1 to 0.6] | 0.2 [0.2 to 0.3]
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 1 | 14 | 5 | 12 | 10
  CD8+-S1 at Month 0-Peru | 0 [0 to 0] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 1 | 33 | 8 | 15 | 14
  CD8+-S1 at Month 0-Total | 0 [0 to 0] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 0 | 19 | 3 | 3 | 4
  CD8+-S1 at Month 0-USA |  | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 3 | 4 | 2 | 4 | 5
  CD8+-S2 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.7 [0.3 to 1.4] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2]
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 4 | 11 | 3 | 5 | 7
  CD8+-S2 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.3 [0.1 to 0.7] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 1 | 7 | 1 | 1 | 2
  CD8+-S2 at Month 0-USA | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 4 | 15 | 5 | 12 | 11
  CD8+-Spike at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 5 | 38 | 8 | 15 | 16
  CD8+-Spike at Month 0-Total | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.2]
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 1 | 23 | 3 | 3 | 5
  CD8+-Spike at Month 0-USA | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 1.1] | 0.2 [0.2 to 0.3] | 0.1 [0.1 to 0.2]

30. Primary Outcome: SARS-CoV-2-specific Memory B Cell Response Magnitude (B Cell) by Region and COVID-19 Severity Among America Cohort
Description: SARS-CoV-2-specific B cell responses and B cell phenotypic data was identified and characterized using fluorescently-labelled recombinant Env proteins (S6P and RBD) in combination with a flow cytometry antibody panel on all available samples from the enrollment visit (V1). The sample will be included in the analysis only if the number of IgD- B cells is equal or greater than 1000 for that sample.
  The table summarized SARS-CoV-2-specific Memory B Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and COVID-19 severity among America Cohort (USA and Peru)
Time Frame: Measured at Months 0
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 86 | 150 | 25 | 76 | 51
percentage of cells
  %RBD+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %RBD+ IgA+ of Memory B Cells-Peru | 0.01 [0 to 0.02] | 0.01 [0 to 0.04] | 0.02 [0 to 0.04] | 0.02 [0 to 0.04] | 0.01 [0 to 0.05]
  %RBD+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %RBD+ IgA+ of Memory B Cells-Total | 0.01 [0 to 0.04] | 0.01 [0 to 0.03] | 0.02 [0 to 0.04] | 0.01 [0 to 0.04] | 0 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %RBD+ IgA+ of Memory B Cells-USA | 0 [0 to 0.04] | 0.01 [0 to 0.02] | 0.02 [0.02 to 0.05] | 0 [0 to 0.05] | 0 [0 to 0.01]
  %RBD+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %RBD+ IgG+ of Memory B Cells-Peru | 0.08 [0.04 to 0.15] | 0.14 [0.06 to 0.3] | 0.13 [0.04 to 0.31] | 0.23 [0.11 to 0.35] | 0.23 [0.13 to 0.36]
  %RBD+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %RBD+ IgG+ of Memory B Cells-Total | 0.09 [0.01 to 0.18] | 0.14 [0.05 to 0.28] | 0.15 [0.08 to 0.31] | 0.25 [0.11 to 0.35] | 0.23 [0.13 to 0.36]
  %RBD+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %RBD+ IgG+ of Memory B Cells-USA | 0.1 [0 to 0.23] | 0.13 [0.05 to 0.25] | 0.24 [0.19 to 0.32] | 0.27 [0.08 to 0.41] | 0.23 [0.1 to 0.38]
  %RBD+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %RBD+ IgM+ of Memory B Cells-Peru | 0 [0 to 0.02] | 0 [0 to 0.02] | 0 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %RBD+ IgM+ of Memory B Cells-Total | 0 [0 to 0.02] | 0 [0 to 0.02] | 0 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0]
  %RBD+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %RBD+ IgM+ of Memory B Cells-USA | 0 [0 to 0.03] | 0 [0 to 0.01] | 0.03 [0 to 0.07] | 0 [0 to 0.02] | 0 [0 to 0]
  %RBD+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %RBD+ of Total B Cells-Peru | 0.05 [0.03 to 0.09] | 0.08 [0.05 to 0.14] | 0.08 [0.05 to 0.11] | 0.1 [0.05 to 0.14] | 0.09 [0.07 to 0.13]
  %RBD+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %RBD+ of Total B Cells-Total | 0.05 [0.03 to 0.12] | 0.06 [0.04 to 0.11] | 0.08 [0.05 to 0.11] | 0.08 [0.05 to 0.14] | 0.07 [0.05 to 0.12]
  %RBD+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %RBD+ of Total B Cells-USA | 0.06 [0.02 to 0.16] | 0.04 [0.03 to 0.07] | 0.08 [0.06 to 0.2] | 0.07 [0.04 to 0.12] | 0.05 [0.02 to 0.07]
  %S+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgA+ of Memory B Cells-Peru | 0.06 [0.03 to 0.09] | 0.08 [0.04 to 0.12] | 0.09 [0.04 to 0.21] | 0.07 [0.03 to 0.15] | 0.08 [0.04 to 0.15]
  %S+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgA+ of Memory B Cells-Total | 0.04 [0.01 to 0.08] | 0.08 [0.03 to 0.12] | 0.07 [0.04 to 0.15] | 0.07 [0.03 to 0.12] | 0.06 [0.02 to 0.1]
  %S+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgA+ of Memory B Cells-USA | 0.04 [0.01 to 0.08] | 0.07 [0.03 to 0.11] | 0.04 [0.04 to 0.07] | 0.07 [0.03 to 0.1] | 0.04 [0 to 0.08]
  %S+ IgA+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgA+ of Total B Cells-Peru | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.06] | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.03]
  %S+ IgA+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgA+ of Total B Cells-Total | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.06] | 0.01 [0.01 to 0.03] | 0.01 [0 to 0.02]
  %S+ IgA+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgA+ of Total B Cells-USA | 0.01 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0 [0 to 0.01]
  %S+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgG+ of Memory B Cells-Peru | 0.39 [0.2 to 0.6] | 0.63 [0.38 to 1.07] | 0.78 [0.32 to 1.32] | 1.02 [0.6 to 1.26] | 1.09 [0.63 to 1.4]
  %S+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgG+ of Memory B Cells-Total | 0.33 [0.07 to 0.61] | 0.63 [0.38 to 1.02] | 0.95 [0.33 to 1.32] | 1.07 [0.55 to 1.43] | 1.08 [0.61 to 1.43]
  %S+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgG+ of Memory B Cells-USA | 0.28 [0.05 to 0.61] | 0.63 [0.36 to 1] | 0.98 [0.75 to 1.38] | 1.13 [0.46 to 1.73] | 1.07 [0.44 to 1.6]
  %S+ IgG+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgG+ of Total B Cells-Peru | 0.07 [0.04 to 0.15] | 0.17 [0.08 to 0.26] | 0.2 [0.12 to 0.26] | 0.2 [0.14 to 0.33] | 0.24 [0.2 to 0.29]
  %S+ IgG+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgG+ of Total B Cells-Total | 0.06 [0.01 to 0.14] | 0.11 [0.06 to 0.23] | 0.2 [0.12 to 0.23] | 0.2 [0.12 to 0.29] | 0.21 [0.1 to 0.26]
  %S+ IgG+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgG+ of Total B Cells-USA | 0.05 [0.01 to 0.14] | 0.1 [0.06 to 0.17] | 0.17 [0.12 to 0.22] | 0.2 [0.11 to 0.25] | 0.16 [0.05 to 0.22]
  %S+ IgM+ IgD+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgM+ IgD+ of Total B Cells-Peru | 0.11 [0.08 to 0.13] | 0.14 [0.1 to 0.18] | 0.11 [0.09 to 0.15] | 0.09 [0.08 to 0.13] | 0.11 [0.08 to 0.14]
  %S+ IgM+ IgD+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgM+ IgD+ of Total B Cells-Total | 0.08 [0.06 to 0.12] | 0.11 [0.08 to 0.16] | 0.1 [0.09 to 0.15] | 0.1 [0.08 to 0.14] | 0.1 [0.06 to 0.14]
  %S+ IgM+ IgD+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgM+ IgD+ of Total B Cells-USA | 0.08 [0.05 to 0.1] | 0.09 [0.07 to 0.12] | 0.1 [0.07 to 0.13] | 0.11 [0.07 to 0.17] | 0.1 [0.06 to 0.14]
  %S+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgM+ of Memory B Cells-Peru | 0.03 [0 to 0.06] | 0.04 [0.02 to 0.09] | 0.04 [0.02 to 0.08] | 0.04 [0.01 to 0.06] | 0.04 [0.02 to 0.09]
  %S+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgM+ of Memory B Cells-Total | 0.03 [0 to 0.07] | 0.05 [0.03 to 0.09] | 0.04 [0.02 to 0.09] | 0.04 [0.01 to 0.06] | 0.03 [0 to 0.07]
  %S+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgM+ of Memory B Cells-USA | 0.03 [0 to 0.07] | 0.06 [0.03 to 0.09] | 0.07 [0.02 to 0.12] | 0.04 [0 to 0.07] | 0.02 [0 to 0.05]
  %S+ IgM+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ IgM+ of Total B Cells-Peru | 0.01 [0 to 0.01] | 0.01 [0.01 to 0.03] | 0.01 [0 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ IgM+ of Total B Cells-Total | 0.01 [0 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.01] | 0 [0 to 0.02]
  %S+ IgM+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ IgM+ of Total B Cells-USA | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.03] | 0 [0 to 0.01] | 0 [0 to 0.01]
  %S+ of Total B Cells-Peru: number analyzed (Participants) | 24 | 49 | 12 | 36 | 25
  %S+ of Total B Cells-Peru | 0.29 [0.16 to 0.37] | 0.43 [0.26 to 0.59] | 0.43 [0.27 to 0.59] | 0.43 [0.32 to 0.55] | 0.43 [0.38 to 0.52]
  %S+ of Total B Cells-Total: number analyzed (Participants) | 62 | 107 | 16 | 62 | 44
  %S+ of Total B Cells-Total | 0.22 [0.12 to 0.33] | 0.31 [0.22 to 0.5] | 0.36 [0.3 to 0.52] | 0.42 [0.29 to 0.55] | 0.4 [0.3 to 0.48]
  %S+ of Total B Cells-USA: number analyzed (Participants) | 38 | 58 | 4 | 26 | 19
  %S+ of Total B Cells-USA | 0.21 [0.1 to 0.32] | 0.26 [0.2 to 0.37] | 0.34 [0.3 to 0.4] | 0.37 [0.27 to 0.54] | 0.3 [0.17 to 0.41]

31. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG1) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2, 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: less than 28 days since SARS-CoV-2 diagnosis
- Group 2: 28-41 days since SARS-CoV-2 diagnosis
- Group 3: 42-55 days since SARS-CoV-2 diagnosis
- Group 4: 56+ days since SARS-CoV-2 diagnosis
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 20 | 63 | 69 | 132
  2019-nCoV S/293F-50 at Month 0-Total | 20 | 60 | 63 | 121
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 22 | 60 | 63 | 127
  2019-nCoV S/293F-50 at Month 2-Total | 21 | 57 | 57 | 115
  2019-nCoV S/293F-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 84
  2019-nCoV S/293F-50 at Month 4-Total | 21 | 45 | 42 | 75
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 30 | 81 | 90 | 166
  SARS-CoV-2 DB His-50 at Month 0-Total | 28 | 72 | 78 | 148
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 63 | 129
  SARS-CoV-2 DB His-50 at Month 2-Total | 22 | 56 | 55 | 114
  SARS-CoV-2 DB His-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 48 | 83
  SARS-CoV-2 DB His-50 at Month 4-Total | 21 | 44 | 40 | 72
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 30 | 81 | 90 | 166
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 28 | 71 | 78 | 147
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 21 | 59 | 64 | 125
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 20 | 54 | 55 | 110
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total: number analyzed (Participants) | 20 | 45 | 45 | 80
  SARS-CoV-2 Nucleoprotein His-50 at Month 4-Total | 20 | 38 | 37 | 69
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 14 | 62 | 65 | 123
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 13 | 58 | 61 | 112
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 66 | 126
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 22 | 56 | 59 | 112
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total: number analyzed (Participants) | 21 | 47 | 49 | 83
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 4-Total | 21 | 44 | 42 | 74
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 27 | 81 | 86 | 164
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 24 | 72 | 77 | 144
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 23 | 61 | 65 | 128
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 22 | 57 | 58 | 112
  SARS-CoV-2 S1 C His-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 48 | 83
  SARS-CoV-2 S1 C His-50 at Month 4-Total | 21 | 44 | 41 | 72
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 30 | 80 | 90 | 165
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 28 | 72 | 82 | 149
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 20 | 58 | 62 | 125
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 19 | 55 | 57 | 115
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 19 | 45 | 42 | 82
  SARS-CoV-2 S1S2 ECD His-50 at Month 4-Total | 19 | 43 | 37 | 73
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 165
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 29 | 74 | 82 | 147
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 66 | 128
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 22 | 56 | 59 | 116
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 84
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 4-Total | 21 | 45 | 42 | 75
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 14 | 63 | 64 | 127
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 14 | 60 | 59 | 114
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 22 | 58 | 65 | 124
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 21 | 54 | 56 | 110
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 83
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 4-Total | 21 | 45 | 42 | 72

32. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG1) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by BAMA IgG1 at Visit 1, 2, 3, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2, 4
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
MFI
  2019-nCoV S/293F-1000 at Month 0-Total: number analyzed (Participants) | 20 | 63 | 69 | 132
  2019-nCoV S/293F-1000 at Month 0-Total | 11484.4 [5568.6 to 20553.6] | 22000 [10672.4 to 22000] | 22000 [5914.2 to 22000] | 14553.4 [4370.4 to 22000]
  2019-nCoV S/293F-1000 at Month 2-Total: number analyzed (Participants) | 22 | 60 | 63 | 127
  2019-nCoV S/293F-1000 at Month 2-Total | 5544.1 [1989.5 to 12245.6] | 11097.6 [3760.7 to 22000] | 9271.5 [1901.1 to 21065] | 8335.5 [2706.8 to 18749.2]
  2019-nCoV S/293F-1000 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 84
  2019-nCoV S/293F-1000 at Month 4-Total | 2156 [951.2 to 4403.2] | 6349 [1452.9 to 19026.9] | 3660 [1538 to 14339] | 3067.9 [978.9 to 10026.9]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 14 | 61 | 65 | 120
  229E-RBD-50 at Month 0-Total | 5759.9 [3973.1 to 8372.8] | 5035.8 [3799.8 to 7984.2] | 5897.8 [3326.8 to 8369.5] | 5698 [3337.4 to 8032.5]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 21 | 59 | 60 | 121
  229E-RBD-50 at Month 2-Total | 6586 [4399 to 8187.2] | 5076 [2771.9 to 7887.1] | 5212.5 [3398.5 to 7946.4] | 4738.2 [2894.5 to 7440]
  229E-RBD-50 at Month 4-Total: number analyzed (Participants) | 20 | 45 | 40 | 76
  229E-RBD-50 at Month 4-Total | 5714 [3953.8 to 8962.4] | 6275.5 [3624 to 8627.8] | 6810.4 [4639.9 to 9987.6] | 6235.8 [3862.9 to 8359.8]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 76 | 86 | 149
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 18341.8 [13014.6 to 22000] | 15357.9 [9446.6 to 21100.9] | 13943.4 [7657.2 to 22000] | 12162.5 [6134.8 to 21400.2]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 21 | 58 | 62 | 122
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 13942 [8989.5 to 17316.2] | 9134.4 [5638.7 to 16769.2] | 8646.8 [5308.2 to 15402.4] | 9715.4 [5260.2 to 14721.7]
  HCoV-229E S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 21 | 47 | 44 | 82
  HCoV-229E S1S2 ECD His-50 at Month 4-Total | 11015.5 [8560.8 to 13422.3] | 9341 [5824.8 to 14489] | 10458.6 [6214.4 to 19640.3] | 10425.4 [5139.8 to 14758.9]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 76 | 86 | 148
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 18176.8 [12582.2 to 22000] | 14720.5 [8018.5 to 21628.1] | 16978.4 [9741.4 to 22000] | 14320 [6958.1 to 22000]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 21 | 58 | 61 | 123
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 17001.8 [10625.8 to 22000] | 16950.5 [9025.9 to 21921.2] | 13674.5 [7867.2 to 20084.5] | 12047.8 [7491.2 to 18459.5]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 48 | 83
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 4-Total | 16352.5 [7446.2 to 20204.3] | 14488 [7171.8 to 20768.1] | 11621.1 [8427.3 to 19273.6] | 12100.8 [6926.9 to 21509.1]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 76 | 85 | 150
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 1310.2 [759.1 to 2238] | 1197.9 [37.8 to 2493.1] | 1319.2 [94 to 3097.5] | 1318.1 [8.6 to 3213.3]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 19 | 53 | 55 | 112
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 2241 [1118.1 to 5181.4] | 1799.2 [602 to 3704.5] | 1653.8 [586.9 to 3214.2] | 1478.9 [371.1 to 4411.1]
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 19 | 47 | 46 | 82
  HCoV-NL63 S1S2 ECD His-50 at Month 4-Total | 2414.3 [1354.6 to 3212] | 1363.5 [858.1 to 2593.1] | 1315.8 [638.5 to 2685.6] | 1513.8 [603.6 to 3079.9]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 76 | 86 | 149
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 22000 [19473.1 to 22000] | 22000 [17385.5 to 22000] | 22000 [19581.8 to 22000] | 21808.2 [16243.2 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 21 | 59 | 62 | 122
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 22000 [22000 to 22000] | 22000 [17780.2 to 22000] | 22000 [17461.8 to 22000] | 21969 [12920 to 22000]
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 46 | 82
  HCoV-OC43 S1S2 ECD His-50 at Month 4-Total | 22000 [14702 to 22000] | 22000 [15984.6 to 22000] | 20646.2 [15675.1 to 22000] | 20511.8 [13061.6 to 22000]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 14 | 63 | 65 | 120
  HKU1-RBD-50 at Month 0-Total | 5172.5 [3086.1 to 7727.9] | 4688 [2801.8 to 6782.4] | 4923.8 [3305.5 to 6598.2] | 4291.9 [2400.6 to 6036.5]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 20 | 57 | 59 | 120
  HKU1-RBD-50 at Month 2-Total | 4731.2 [3587.2 to 5942.7] | 4175 [1724.5 to 6107] | 4311.8 [2721.6 to 6346.9] | 3500.8 [1722.1 to 5579.1]
  HKU1-RBD-50 at Month 4-Total: number analyzed (Participants) | 18 | 40 | 41 | 77
  HKU1-RBD-50 at Month 4-Total | 5317.8 [3437.4 to 8881.1] | 5189.4 [3668.8 to 6956.1] | 5507.8 [3667.8 to 8611.8] | 5373 [2680.8 to 7775]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 14 | 63 | 65 | 121
  NL63-RBD-50 at Month 0-Total | 14352.5 [10012.1 to 17704] | 12258.5 [9916.6 to 14972.5] | 10779.8 [8010.2 to 16454.8] | 11885.5 [8681.8 to 15936.8]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 21 | 59 | 62 | 123
  NL63-RBD-50 at Month 2-Total | 16886.5 [15225 to 20130.5] | 15328.8 [10445.8 to 18107.5] | 14236.9 [9743.9 to 18173.8] | 13644.5 [9569.6 to 18060.5]
  NL63-RBD-50 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 46 | 84
  NL63-RBD-50 at Month 4-Total | 16381 [13413.5 to 20575.2] | 15586.1 [12530.4 to 18276.2] | 16318.5 [13572.4 to 19782.6] | 16580.9 [12363.9 to 19943.2]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 14 | 63 | 65 | 118
  OC43-RBD-50 at Month 0-Total | 5351.5 [2714.1 to 8942] | 4108.8 [2664 to 6770] | 4605 [1951.8 to 8643.8] | 3927.1 [2424 to 6054.8]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 21 | 57 | 60 | 121
  OC43-RBD-50 at Month 2-Total | 6109.2 [3276.5 to 10408.5] | 4069.5 [2011.8 to 6808] | 4491.9 [2332.1 to 7179.9] | 4055.2 [2286 to 6998]
  OC43-RBD-50 at Month 4-Total: number analyzed (Participants) | 19 | 43 | 40 | 79
  OC43-RBD-50 at Month 4-Total | 4053.5 [2698 to 9458.4] | 5068.2 [2519.1 to 7666.6] | 5437 [3126.5 to 9777.9] | 5267.5 [2268 to 7898.2]
  SARS-CoV-2 DB His-1000 at Month 0-Total: number analyzed (Participants) | 30 | 81 | 90 | 166
  SARS-CoV-2 DB His-1000 at Month 0-Total | 3903.4 [1181.2 to 8940] | 8110.5 [1056 to 21923.8] | 6366.4 [988.6 to 21668.6] | 4628.9 [1459.1 to 13579.6]
  SARS-CoV-2 DB His-1000 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 63 | 129
  SARS-CoV-2 DB His-1000 at Month 2-Total | 1660.8 [683.6 to 2666.8] | 2814.6 [587.9 to 10179.6] | 1729.8 [355.6 to 8003.2] | 1609 [499.8 to 4622.8]
  SARS-CoV-2 DB His-1000 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 48 | 83
  SARS-CoV-2 DB His-1000 at Month 4-Total | 463.5 [279.2 to 1194] | 1509.5 [310.9 to 5133.3] | 1116.8 [324.4 to 4087.5] | 853.5 [274.5 to 2743.8]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total: number analyzed (Participants) | 30 | 81 | 90 | 166
  SARS-CoV-2 Nucleoprotein His-1000 at Month 0-Total | 2736.9 [1040.4 to 19813.4] | 13506.2 [2016.5 to 22000] | 13011.4 [1628.9 to 22000] | 12524.4 [2197.4 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total: number analyzed (Participants) | 21 | 59 | 64 | 125
  SARS-CoV-2 Nucleoprotein His-1000 at Month 2-Total | 808.5 [587.8 to 5196] | 2651.8 [751.1 to 6471.6] | 2231.6 [386 to 8176.2] | 2878 [603.8 to 8151.2]
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total: number analyzed (Participants) | 20 | 45 | 45 | 80
  SARS-CoV-2 Nucleoprotein His-1000 at Month 4-Total | 321.1 [167.5 to 1147.1] | 760.8 [240.2 to 2111] | 509.2 [242.5 to 2733] | 556.9 [236.8 to 1680]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total: number analyzed (Participants) | 14 | 62 | 65 | 123
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 0-Total | 2008.6 [935.9 to 4564.1] | 9659.2 [1642.7 to 21640.7] | 9512.8 [1148 to 17840.2] | 3997.5 [1077.9 to 11198.4]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 66 | 126
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 2-Total | 1337.2 [559.6 to 3004.9] | 2169.6 [639.9 to 8637.3] | 1999.5 [304.2 to 7686.8] | 1759.8 [499.2 to 4893.2]
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total: number analyzed (Participants) | 21 | 47 | 49 | 83
  SARS-CoV-2 S Hexapro_293F_PPF-1000 at Month 4-Total | 511.2 [284.5 to 978.2] | 1627 [312.2 to 5317.2] | 834.2 [335.8 to 4397.5] | 636.5 [201.9 to 2993.8]
  SARS-CoV-2 S1 C His-1000 at Month 0-Total: number analyzed (Participants) | 27 | 81 | 86 | 164
  SARS-CoV-2 S1 C His-1000 at Month 0-Total | 3073.5 [1047.4 to 8787.6] | 7604.5 [596.2 to 22000] | 5603.8 [718.8 to 21419.6] | 3894.1 [1204.7 to 14907.9]
  SARS-CoV-2 S1 C His-1000 at Month 2-Total: number analyzed (Participants) | 23 | 61 | 65 | 128
  SARS-CoV-2 S1 C His-1000 at Month 2-Total | 1460.2 [355.9 to 2154.8] | 2109.2 [368.8 to 10737.2] | 1499 [226.2 to 6875.8] | 1481.8 [265.2 to 5454.8]
  SARS-CoV-2 S1 C His-1000 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 48 | 83
  SARS-CoV-2 S1 C His-1000 at Month 4-Total | 427 [195.5 to 1025.5] | 1459.6 [236.2 to 5309.6] | 741.9 [232.6 to 4402.1] | 771.2 [190.1 to 2820.1]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total: number analyzed (Participants) | 30 | 80 | 90 | 165
  SARS-CoV-2 S1S2 ECD His-1000 at Month 0-Total | 3146.6 [972.2 to 5793.9] | 4770.2 [1143.1 to 20761.3] | 7640.1 [1228.6 to 15861.9] | 5985 [1353.8 to 12621]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total: number analyzed (Participants) | 20 | 58 | 62 | 125
  SARS-CoV-2 S1S2 ECD His-1000 at Month 2-Total | 1136.9 [675.5 to 2609.5] | 2766.2 [620.3 to 9405] | 2739.5 [316.5 to 8066.1] | 2470 [555.2 to 7924.2]
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total: number analyzed (Participants) | 19 | 45 | 42 | 82
  SARS-CoV-2 S1S2 ECD His-1000 at Month 4-Total | 701 [381.5 to 968.1] | 2099.2 [365.8 to 6293.5] | 1144.4 [254.6 to 5062.8] | 923.2 [179.9 to 4231.8]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 165
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 0-Total | 9507.8 [4309 to 16696.6] | 19343.6 [5322.3 to 22000] | 14710.5 [6038 to 22000] | 13203.8 [5043.8 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total: number analyzed (Participants) | 23 | 60 | 66 | 128
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 2-Total | 4872.2 [2458.5 to 10428.5] | 9217.9 [3680.4 to 22000] | 8247.1 [1888.5 to 19664.8] | 7916.5 [2783.6 to 17910.9]
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 84
  SARS-CoV-2 spike (PreS Nexelis)-1000 at Month 4-Total | 2363.7 [1155 to 3935.8] | 7105 [1642.2 to 16111.9] | 3783 [1509.8 to 13837.2] | 2925.1 [1103.9 to 10373.2]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total: number analyzed (Participants) | 14 | 63 | 64 | 127
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 0-Total | 1747 [293.9 to 3858.4] | 12005 [1362.6 to 22000] | 8313.6 [845.2 to 22000] | 3940.2 [404.1 to 13471.5]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total: number analyzed (Participants) | 22 | 58 | 65 | 124
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 2-Total | 415.4 [91.3 to 1434.9] | 1863.6 [117.6 to 7913.3] | 685.2 [60.8 to 8406.5] | 872.1 [114.8 to 3358.4]
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total: number analyzed (Participants) | 21 | 48 | 49 | 83
  SARS-CoV-2-NTD-AVI Biotin-1000 at Month 4-Total | 96.3 [24.5 to 567.8] | 512 [94.3 to 3209.9] | 332 [26.5 to 2540.2] | 279.2 [27.8 to 1415.2]

33. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG3) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 89 | 168
  2019-nCoV S/293F-50 at Month 0-Total | 29 | 73 | 77 | 151
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  2019-nCoV S/293F-50 at Month 2-Total | 1 | 19 | 22 | 41
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 89 | 168
  SARS-CoV-2 DB His-50 at Month 0-Total | 26 | 63 | 70 | 136
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 DB His-50 at Month 2-Total | 1 | 10 | 14 | 20
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 89 | 167
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 31 | 75 | 79 | 150
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 1 | 19 | 23 | 33
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 30 | 82 | 87 | 168
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 26 | 65 | 72 | 140
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 1 | 10 | 14 | 32
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 90 | 168
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 27 | 65 | 74 | 141
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 1 | 11 | 16 | 32
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 90 | 166
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 28 | 73 | 78 | 154
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 1 | 21 | 24 | 43
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 90 | 168
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 29 | 74 | 78 | 150
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 1 | 17 | 21 | 41
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 89 | 168
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 28 | 66 | 73 | 143
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 1 | 17 | 19 | 39

34. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG3) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
MFI
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 89 | 168
  2019-nCoV S/293F-50 at Month 0-Total | 5275.2 [3138.2 to 10723.5] | 7354.2 [2928 to 13468.5] | 6335.5 [3196 to 12738] | 6180.5 [3182.8 to 11493.4]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  2019-nCoV S/293F-50 at Month 2-Total | 3674 [3674 to 3674] | 2815.5 [738.2 to 4352.5] | 1935.5 [447.2 to 4011] | 3562 [1412.5 to 6152.2]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 29 | 79 | 89 | 161
  229E-RBD-50 at Month 0-Total | 343 [97 to 460.5] | 210.2 [9.9 to 386.4] | 242.2 [72.2 to 531] | 230.8 [31.5 to 490.2]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 28 | 49
  229E-RBD-50 at Month 2-Total | 47 [47 to 47] | 1 [1 to 6] | 1 [1 to 155.9] | 1 [1 to 1]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 80 | 90 | 168
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 61.8 [1 to 147] | 11.1 [1 to 70.7] | 15.4 [1 to 116.3] | 1 [1 to 72.3]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 630.2 [630.2 to 630.2] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 79 | 90 | 167
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 321 [124.9 to 754.5] | 296.2 [109.2 to 1192.2] | 302.8 [114 to 598.9] | 557.2 [145 to 1748]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 406.8 [406.8 to 406.8] | 192.5 [1 to 1158.2] | 63 [1 to 326.8] | 306.5 [35.8 to 1225.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 80 | 90 | 168
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 22.2 [1 to 113.5] | 1 [1 to 24.1] | 1 [1 to 70] | 1 [1 to 43.6]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 80 | 90 | 167
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 679 [309.5 to 1903.1] | 519.5 [106.9 to 2237.7] | 380.9 [93.4 to 1072.4] | 555.5 [130.5 to 2408.8]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 28 | 48
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 577.5 [577.5 to 577.5] | 32.2 [1 to 644] | 1 [1 to 260.2] | 1 [1 to 1058.1]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 31 | 78 | 89 | 164
  HKU1-RBD-50 at Month 0-Total | 217 [109.4 to 398.8] | 182.6 [21.9 to 316.9] | 201.5 [75 to 430.5] | 195.9 [22.9 to 410.2]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HKU1-RBD-50 at Month 2-Total | 204 [204 to 204] | 1 [1 to 92.8] | 1 [1 to 103] | 1 [1 to 18]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 27 | 72 | 85 | 162
  NL63-RBD-50 at Month 0-Total | 215.2 [19.2 to 458.5] | 273.5 [92.7 to 416.7] | 200.8 [24.2 to 484.5] | 193.5 [1 to 412.8]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  NL63-RBD-50 at Month 2-Total | 152.5 [152.5 to 152.5] | 1 [1 to 1] | 1 [1 to 81.8] | 1 [1 to 11.2]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 31 | 78 | 88 | 167
  OC43-RBD-50 at Month 0-Total | 218.2 [76 to 369] | 157.9 [5.8 to 278.3] | 145.2 [16.5 to 341.9] | 124 [1 to 409.4]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  OC43-RBD-50 at Month 2-Total | 50.5 [50.5 to 50.5] | 1 [1 to 1] | 1 [1 to 48.5] | 1 [1 to 28.8]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 89 | 168
  SARS-CoV-2 DB His-50 at Month 0-Total | 1962.5 [556.9 to 3298.5] | 2412.8 [474.8 to 4158.2] | 1581.2 [709.2 to 3565.5] | 1700 [642.9 to 3822.1]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 DB His-50 at Month 2-Total | 1393.8 [1393.8 to 1393.8] | 406.2 [19.5 to 1083] | 171.2 [1 to 918.2] | 205.8 [1 to 974.2]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 89 | 167
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 6657.2 [3747.1 to 14044.9] | 8643.2 [4124.6 to 17004.2] | 7041 [2795.5 to 11746.8] | 7569.5 [3027.1 to 14175.5]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 1482.5 [1482.5 to 1482.5] | 2162.8 [789 to 7057.8] | 2270 [442.2 to 3598.2] | 1330.8 [246 to 3523.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 30 | 82 | 87 | 168
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 1908.4 [582.6 to 3257.1] | 1739.8 [484.5 to 4570.2] | 1538 [531.6 to 4306.8] | 1670.5 [540.8 to 4214.4]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 790 [790 to 790] | 192.5 [45.2 to 1028.8] | 210.8 [1 to 926] | 565 [36 to 1088.8]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 90 | 168
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 1233.2 [494.2 to 2949] | 2218.9 [358.8 to 5177.3] | 1769.9 [524.5 to 4168.4] | 1702.4 [666.5 to 3998.9]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 1479.5 [1479.5 to 1479.5] | 414.2 [16 to 1515.5] | 290.5 [1 to 1200.5] | 662 [127.8 to 1313.2]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 90 | 166
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 7638.2 [4298.5 to 15088.2] | 9566.2 [3286.8 to 21444.8] | 7286.5 [3736.6 to 19084.7] | 8632.8 [4030.4 to 18051.4]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 2903.8 [2903.8 to 2903.8] | 5407.5 [2462.2 to 8652.2] | 3503.5 [1660.2 to 9682.5] | 4610 [2062 to 11666.2]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 90 | 168
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 4576.5 [2270.9 to 7342] | 5373.1 [1932.1 to 8753.1] | 4580.9 [2000.5 to 8407.5] | 4309.1 [2349.2 to 8847.6]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 2345.2 [2345.2 to 2345.2] | 2048 [539 to 2600.5] | 1415.2 [377 to 2429.5] | 2385.5 [946 to 3879]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 89 | 168
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 1529 [438.1 to 7685.1] | 3675.8 [431.4 to 11368.1] | 2504.8 [394.8 to 6504.2] | 2839.1 [641.9 to 7226.2]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 1487.2 [1487.2 to 1487.2] | 603.2 [144.8 to 974] | 207.5 [1 to 999] | 844 [145 to 1905.5]

35. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgA) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: 28 - 41 days since SARS-CoV-2 diagnosis
- Group 3: 42 - 55 days since SARS-CoV-2 diagnosis
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  2019-nCoV S/293F-50 at Month 0-Total | 29 | 74 | 80 | 146
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  2019-nCoV S/293F-50 at Month 2-Total | 1 | 18 | 24 | 43
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 DB His-50 at Month 0-Total | 24 | 66 | 69 | 124
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 DB His-50 at Month 2-Total | 0 | 15 | 19 | 31
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 28 | 75 | 77 | 142
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 0 | 20 | 20 | 39
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 29 | 74 | 81 | 149
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 1 | 19 | 26 | 42
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 29 | 71 | 76 | 146
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 1 | 17 | 23 | 40
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 12 | 42 | 40 | 74
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 0 | 6 | 8 | 17
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 29 | 70 | 78 | 138
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 1 | 16 | 21 | 41
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 20 | 64 | 69 | 122
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 14 | 53 | 49 | 91
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 0 | 15 | 16 | 29

36. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgA) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
MFI
  2019-nCoV S/293F-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  2019-nCoV S/293F-50 at Month 0-Total | 8344.8 [2822.9 to 16328.2] | 8379.1 [3444.2 to 18318.1] | 8258.5 [3107.2 to 15027.2] | 5754.8 [2256 to 10838]
  2019-nCoV S/293F-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  2019-nCoV S/293F-50 at Month 2-Total | 11670.8 [11670.8 to 11670.8] | 4340.5 [1324.5 to 7052] | 3227.5 [1887 to 7967.5] | 2781.2 [1566.5 to 6886.2]
  229E-RBD-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  229E-RBD-50 at Month 0-Total | 481.5 [354.4 to 833.4] | 585.4 [330.9 to 904.4] | 625.5 [294.6 to 1097.2] | 459.5 [283.8 to 886]
  229E-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  229E-RBD-50 at Month 2-Total | 299.2 [299.2 to 299.2] | 250.2 [204.2 to 382.2] | 306.2 [202.8 to 480.5] | 508.8 [282.8 to 909.8]
  HCoV-229E S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  HCoV-229E S1S2 ECD His-50 at Month 0-Total | 508.8 [281 to 1276] | 422.6 [233.3 to 882.8] | 465.8 [278.6 to 1014.8] | 450 [190.8 to 932.5]
  HCoV-229E S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-229E S1S2 ECD His-50 at Month 2-Total | 278.2 [278.2 to 278.2] | 387 [258.8 to 698] | 575.2 [171 to 918.5] | 614.2 [176 to 1250.2]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 0-Total | 791.2 [544.1 to 2471.5] | 1293.8 [579.1 to 2530.2] | 1414.2 [660.6 to 3152.2] | 1510.5 [671 to 3996.8]
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-HKU1 N5 S1S2 ECD His-50 at Month 2-Total | 2649.2 [2649.2 to 2649.2] | 947 [589 to 1494] | 1010 [471 to 2905.5] | 1714.2 [756.5 to 4510.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  HCoV-NL63 S1S2 ECD His-50 at Month 0-Total | 73.2 [23.6 to 174.2] | 74.1 [18.9 to 180] | 89.2 [28.8 to 199.9] | 86.5 [39 to 196.2]
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 47
  HCoV-NL63 S1S2 ECD His-50 at Month 2-Total | 251.2 [251.2 to 251.2] | 49.5 [18.2 to 219.5] | 90.8 [50.2 to 165.2] | 92 [61.4 to 165.6]
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  HCoV-OC43 S1S2 ECD His-50 at Month 0-Total | 2960.5 [1315.6 to 4959.8] | 3252.2 [1508.9 to 5773.4] | 2649 [1489.4 to 6131.1] | 3493 [1618 to 7392.2]
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HCoV-OC43 S1S2 ECD His-50 at Month 2-Total | 4475.8 [4475.8 to 4475.8] | 1773.8 [866.8 to 3461.5] | 2548 [1159.5 to 4868.8] | 3401.2 [1486.2 to 7176.2]
  HKU1-RBD-50 at Month 0-Total: number analyzed (Participants) | 30 | 82 | 91 | 169
  HKU1-RBD-50 at Month 0-Total | 515.5 [268.2 to 712.2] | 448 [288.6 to 847.8] | 490.2 [287 to 832.5] | 436.8 [281.5 to 842.5]
  HKU1-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  HKU1-RBD-50 at Month 2-Total | 293.5 [293.5 to 293.5] | 358.2 [181.5 to 774.5] | 376.2 [210.8 to 559.5] | 447.8 [236 to 847]
  NL63-RBD-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  NL63-RBD-50 at Month 0-Total | 1086.5 [805.5 to 1795.9] | 1097.6 [697.4 to 2026.8] | 1582.5 [849 to 2724.6] | 1166.5 [596.2 to 2984]
  NL63-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  NL63-RBD-50 at Month 2-Total | 604 [604 to 604] | 774.8 [637.8 to 1646.5] | 1395.8 [689 to 2225.5] | 1269.5 [676 to 3253.5]
  OC43-RBD-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  OC43-RBD-50 at Month 0-Total | 463.8 [229 to 919.1] | 486 [305.1 to 965.7] | 431.5 [294.4 to 1076.5] | 547 [289.8 to 1032.8]
  OC43-RBD-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  OC43-RBD-50 at Month 2-Total | 245 [245 to 245] | 299 [225.2 to 668.8] | 477.8 [250 to 821.2] | 708.8 [293.5 to 1571.5]
  SARS-CoV-2 DB His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 DB His-50 at Month 0-Total | 3886.2 [1076.9 to 8525.4] | 4630.8 [1414.1 to 9779.6] | 3334 [893.9 to 7987.5] | 2041.2 [730.8 to 5161]
  SARS-CoV-2 DB His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 DB His-50 at Month 2-Total | 630.8 [630.8 to 630.8] | 1916.8 [814.2 to 3611.5] | 1949.8 [469 to 4851.2] | 1634.5 [509.8 to 3837.5]
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 Nucleoprotein His-50 at Month 0-Total | 2037.2 [765.6 to 4656.2] | 3927.8 [759.2 to 7898.6] | 2168.5 [531.6 to 6033.9] | 1297.8 [489.8 to 3912.8]
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 Nucleoprotein His-50 at Month 2-Total | 209.2 [209.2 to 209.2] | 849.2 [431.2 to 1566.2] | 641.8 [278.8 to 1748.2] | 908.2 [434 to 2736.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 0-Total | 3866.8 [1276.2 to 8121.1] | 3721.9 [1385.1 to 10293.8] | 3279.5 [981.9 to 7809.2] | 2026.5 [833.5 to 5152.5]
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50 at Month 2-Total | 3622.8 [3622.8 to 3622.8] | 1977.2 [593 to 3498.2] | 1578.8 [587.8 to 3617.2] | 1245.8 [817.5 to 2715.8]
  SARS-CoV-2 S1 C His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S1 C His-50 at Month 0-Total | 3496.8 [705.1 to 7280.5] | 3516.6 [965.5 to 10406.3] | 3014.5 [670.2 to 7256.9] | 1579.5 [485 to 4205]
  SARS-CoV-2 S1 C His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1 C His-50 at Month 2-Total | 342.8 [342.8 to 342.8] | 1005.5 [429.5 to 2490] | 760.5 [244.5 to 2695] | 692 [248.8 to 1840.8]
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 S1S2 ECD His-50 at Month 0-Total | 4231.8 [1408.6 to 6416.8] | 5244.9 [1482.2 to 10255.1] | 3988.2 [1884.5 to 7836.8] | 3924.5 [1327.5 to 6737.2]
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 S1S2 ECD His-50 at Month 2-Total | 4205.5 [4205.5 to 4205.5] | 4024.8 [2184.5 to 4734.8] | 3322.5 [1349.2 to 4748.8] | 3798.2 [1901.5 to 5377.8]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total: number analyzed (Participants) | 31 | 82 | 91 | 169
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 0-Total | 7566.2 [2356.5 to 11938.8] | 7185.2 [2694.5 to 14374.1] | 6511.5 [2184 to 12132.6] | 4671.5 [1874 to 10204.2]
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2 spike (PreS Nexelis)-50 at Month 2-Total | 12725.2 [12725.2 to 12725.2] | 3087.5 [1271.8 to 6934.5] | 3058.8 [1070.5 to 8905.5] | 2807 [1846.2 to 5988.8]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total: number analyzed (Participants) | 20 | 64 | 69 | 122
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 0-Total | 1366.9 [216.4 to 6557.6] | 2209.1 [514.8 to 7444.3] | 1690.8 [124 to 5796.5] | 1249.5 [246.5 to 3262.5]
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total: number analyzed (Participants) | 1 | 21 | 29 | 49
  SARS-CoV-2-NTD-AVI Biotin-50 at Month 2-Total | 214.8 [214.8 to 214.8] | 579.8 [176.2 to 2509] | 256.8 [113.2 to 681.8] | 342 [139.8 to 1390]

37. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  VRC7480_G614 at Month 0-Peru: number analyzed (Participants) | 22 | 50 | 52 | 53
  VRC7480_G614 at Month 0-Peru | 21 | 48 | 48 | 50
  VRC7480_G614 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 91 | 168
  VRC7480_G614 at Month 0-Total | 29 | 75 | 80 | 151
  VRC7480_G614 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 39 | 115
  VRC7480_G614 at Month 0-USA | 8 | 27 | 32 | 101
  VRC7480_G614 at Month 12-Peru: number analyzed (Participants) | 0 | 1 | 1 | 5
  VRC7480_G614 at Month 12-Peru |  | 1 | 1 | 5
  VRC7480_G614 at Month 12-Total: number analyzed (Participants) | 1 | 5 | 3 | 14
  VRC7480_G614 at Month 12-Total | 1 | 4 | 3 | 14
  VRC7480_G614 at Month 12-USA: number analyzed (Participants) | 1 | 4 | 2 | 9
  VRC7480_G614 at Month 12-USA | 1 | 3 | 2 | 9
  VRC7480_G614 at Month 2-Peru: number analyzed (Participants) | 16 | 34 | 31 | 25
  VRC7480_G614 at Month 2-Peru | 15 | 31 | 25 | 23
  VRC7480_G614 at Month 2-Total: number analyzed (Participants) | 19 | 53 | 53 | 91
  VRC7480_G614 at Month 2-Total | 18 | 48 | 43 | 82
  VRC7480_G614 at Month 2-USA: number analyzed (Participants) | 3 | 19 | 22 | 66
  VRC7480_G614 at Month 2-USA | 3 | 17 | 18 | 59
  VRC7480_G614 at Month 4-Peru: number analyzed (Participants) | 1 | 1 | 1 | 6
  VRC7480_G614 at Month 4-Peru | 1 | 1 | 1 | 6
  VRC7480_G614 at Month 4-Total: number analyzed (Participants) | 2 | 5 | 2 | 15
  VRC7480_G614 at Month 4-Total | 2 | 5 | 2 | 13
  VRC7480_G614 at Month 4-USA: number analyzed (Participants) | 1 | 4 | 1 | 9
  VRC7480_G614 at Month 4-USA | 1 | 4 | 1 | 7

38. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2,3, 4, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Titer
  VRC7480_G614-ID50 at Month 0-Peru: number analyzed (Participants) | 22 | 50 | 52 | 53
  VRC7480_G614-ID50 at Month 0-Peru | 636.7 [214.7 to 1804.3] | 2322 [631.8 to 5904.3] | 1264 [288.5 to 5638.2] | 574.8 [180 to 1623.6]
  VRC7480_G614-ID50 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 91 | 168
  VRC7480_G614-ID50 at Month 0-Total | 370.7 [155.8 to 931.7] | 1019 [81.8 to 4617.1] | 682.8 [87.1 to 1844.6] | 374.2 [103.2 to 1205]
  VRC7480_G614-ID50 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 39 | 115
  VRC7480_G614-ID50 at Month 0-USA | 216.0 [87.6 to 463] | 71.50 [21.3 to 282.9] | 164.7 [26.4 to 711.4] | 311.5 [76.9 to 1095.6]
  VRC7480_G614-ID50 at Month 12-Peru: number analyzed (Participants) | 0 | 1 | 1 | 5
  VRC7480_G614-ID50 at Month 12-Peru |  | 964.4 [964.4 to 964.4] | 866.7 [866.7 to 866.7] | 120.2 [65.1 to 289.6]
  VRC7480_G614-ID50 at Month 12-Total: number analyzed (Participants) | 1 | 5 | 3 | 14
  VRC7480_G614-ID50 at Month 12-Total | 346.4 [346.4 to 346.4] | 117.8 [94.3 to 281.8] | 707.2 [469.7 to 787] | 267.6 [77.2 to 475.9]
  VRC7480_G614-ID50 at Month 12-USA: number analyzed (Participants) | 1 | 4 | 2 | 9
  VRC7480_G614-ID50 at Month 12-USA | 346.4 [346.4 to 346.4] | 106.1 [72 to 158.8] | 469.7 [351 to 588.5] | 411.9 [113.2 to 608.8]
  VRC7480_G614-ID50 at Month 2-Peru: number analyzed (Participants) | 16 | 34 | 31 | 25
  VRC7480_G614-ID50 at Month 2-Peru | 47.20 [20.6 to 82] | 228.8 [104 to 893.6] | 152.2 [22.6 to 500.1] | 220.7 [47.5 to 347.1]
  VRC7480_G614-ID50 at Month 2-Total: number analyzed (Participants) | 19 | 53 | 53 | 91
  VRC7480_G614-ID50 at Month 2-Total | 51.30 [27.3 to 143.8] | 195.6 [49.1 to 707.2] | 103.5 [35.1 to 356] | 151.7 [44.9 to 380.5]
  VRC7480_G614-ID50 at Month 2-USA: number analyzed (Participants) | 3 | 19 | 22 | 66
  VRC7480_G614-ID50 at Month 2-USA | 151.8 [138.6 to 291.1] | 50.60 [27.2 to 180.2] | 75.00 [36.3 to 156.7] | 120.4 [40.9 to 391.7]
  VRC7480_G614-ID50 at Month 4-Peru: number analyzed (Participants) | 1 | 1 | 1 | 6
  VRC7480_G614-ID50 at Month 4-Peru | 113.2 [113.2 to 113.2] | 151.7 [151.7 to 151.7] | 29.40 [29.4 to 29.4] | 239.0 [121.6 to 370.4]
  VRC7480_G614-ID50 at Month 4-Total: number analyzed (Participants) | 2 | 5 | 2 | 15
  VRC7480_G614-ID50 at Month 4-Total | 183.2 [148.2 to 218.3] | 120.2 [117.8 to 151.7] | 61.90 [45.6 to 78.1] | 281.8 [135.9 to 448.9]
  VRC7480_G614-ID50 at Month 4-USA: number analyzed (Participants) | 1 | 4 | 1 | 9
  VRC7480_G614-ID50 at Month 4-USA | 253.3 [253.3 to 253.3] | 119.0 [103.1 to 271.7] | 94.30 [94.3 to 94.3] | 346.4 [187.1 to 450.2]
  VRC7480_G614-ID80 at Month 0-Peru: number analyzed (Participants) | 22 | 50 | 52 | 53
  VRC7480_G614-ID80 at Month 0-Peru | 129.4 [52.3 to 237.6] | 579.7 [136.6 to 1006.3] | 228.1 [75.3 to 877.2] | 137.2 [56.1 to 364.7]
  VRC7480_G614-ID80 at Month 0-Total: number analyzed (Participants) | 31 | 81 | 91 | 168
  VRC7480_G614-ID80 at Month 0-Total | 120.2 [40.2 to 178.1] | 213.3 [25.5 to 810.2] | 144.0 [29.2 to 554.4] | 105.7 [31.3 to 242]
  VRC7480_G614-ID80 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 39 | 115
  VRC7480_G614-ID80 at Month 0-USA | 54.50 [29.1 to 129.7] | 23.90 [10 to 97.9] | 36.60 [10 to 148.4] | 90.40 [27.1 to 206.8]
  VRC7480_G614-ID80 at Month 12-Peru: number analyzed (Participants) | 0 | 1 | 1 | 5
  VRC7480_G614-ID80 at Month 12-Peru |  | 387.4 [387.4 to 387.4] | 259.2 [259.2 to 259.2] | 46.60 [46.1 to 104.3]
  VRC7480_G614-ID80 at Month 12-Total: number analyzed (Participants) | 1 | 5 | 3 | 14
  VRC7480_G614-ID80 at Month 12-Total | 120.4 [120.4 to 120.4] | 44.10 [30.6 to 111.5] | 189.4 [138.4 to 224.3] | 88.90 [39.5 to 152.7]
  VRC7480_G614-ID80 at Month 12-USA: number analyzed (Participants) | 1 | 4 | 2 | 9
  VRC7480_G614-ID80 at Month 12-USA | 120.4 [120.4 to 120.4] | 37.40 [24.2 to 60.9] | 138.4 [112.9 to 163.9] | 128.3 [37.3 to 182.2]
  VRC7480_G614-ID80 at Month 2-Peru: number analyzed (Participants) | 16 | 34 | 31 | 25
  VRC7480_G614-ID80 at Month 2-Peru | 21.50 [10 to 31.8] | 70.30 [33.1 to 191.2] | 39.40 [10 to 146.1] | 77.40 [25.6 to 135.4]
  VRC7480_G614-ID80 at Month 2-Total: number analyzed (Participants) | 19 | 53 | 53 | 91
  VRC7480_G614-ID80 at Month 2-Total | 24.00 [10 to 45.9] | 51.60 [20.5 to 176.9] | 35.00 [10 to 119.4] | 41.70 [10 to 138.5]
  VRC7480_G614-ID80 at Month 2-USA: number analyzed (Participants) | 3 | 19 | 22 | 66
  VRC7480_G614-ID80 at Month 2-USA | 50.30 [44.4 to 89.3] | 20.50 [10 to 49.6] | 26.90 [10 to 46.7] | 37.50 [10 to 139.4]
  VRC7480_G614-ID80 at Month 4-Peru: number analyzed (Participants) | 1 | 1 | 1 | 6
  VRC7480_G614-ID80 at Month 4-Peru | 37.30 [37.3 to 37.3] | 55.70 [55.7 to 55.7] | 13.70 [13.7 to 13.7] | 80.40 [41.4 to 140.7]
  VRC7480_G614-ID80 at Month 4-Total: number analyzed (Participants) | 2 | 5 | 2 | 15
  VRC7480_G614-ID80 at Month 4-Total | 59.00 [48.1 to 69.8] | 46.60 [44.1 to 55.7] | 22.20 [17.9 to 26.4] | 111.5 [46.6 to 148.4]
  VRC7480_G614-ID80 at Month 4-USA: number analyzed (Participants) | 1 | 4 | 1 | 9
  VRC7480_G614-ID80 at Month 4-USA | 80.70 [80.7 to 80.7] | 45.40 [39.2 to 81.4] | 30.60 [30.6 to 30.6] | 120.4 [62.6 to 138.2]

39. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Days Since SARS-CoV-2 Diagnosis Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and days since SARS-CoV-2 diagnosis group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 83 | 76 | 161
Participants
  SARS-Cov-2 D614G at Month 0-RSA: number analyzed (Participants) | 22 | 51 | 54 | 109
  SARS-Cov-2 D614G at Month 0-RSA | 20 | 48 | 50 | 101
  SARS-Cov-2 D614G at Month 0-Total: number analyzed (Participants) | 24 | 68 | 71 | 157
  SARS-Cov-2 D614G at Month 0-Total | 22 | 61 | 60 | 146
  SARS-Cov-2 D614G at Month 0-non-RSA: number analyzed (Participants) | 2 | 17 | 17 | 48
  SARS-Cov-2 D614G at Month 0-non-RSA | 2 | 13 | 10 | 45
  SARS-Cov-2 D614G at Month 12-RSA: number analyzed (Participants) | 7 | 22 | 24 | 58
  SARS-Cov-2 D614G at Month 12-RSA | 7 | 22 | 24 | 56
  SARS-Cov-2 D614G at Month 12-Total: number analyzed (Participants) | 9 | 34 | 38 | 99
  SARS-Cov-2 D614G at Month 12-Total | 9 | 33 | 37 | 96
  SARS-Cov-2 D614G at Month 12-non-RSA: number analyzed (Participants) | 2 | 12 | 14 | 41
  SARS-Cov-2 D614G at Month 12-non-RSA | 2 | 11 | 13 | 40
  SARS-Cov-2 D614G at Month 2-RSA: number analyzed (Participants) | 16 | 31 | 40 | 70
  SARS-Cov-2 D614G at Month 2-RSA | 15 | 29 | 40 | 63
  SARS-Cov-2 D614G at Month 2-Total: number analyzed (Participants) | 18 | 44 | 56 | 118
  SARS-Cov-2 D614G at Month 2-Total | 16 | 37 | 52 | 106
  SARS-Cov-2 D614G at Month 2-non-RSA: number analyzed (Participants) | 2 | 13 | 16 | 48
  SARS-Cov-2 D614G at Month 2-non-RSA | 1 | 8 | 12 | 43
  SARS-Cov-2 D614G at Month 4-RSA: number analyzed (Participants) | 16 | 31 | 37 | 72
  SARS-Cov-2 D614G at Month 4-RSA | 15 | 27 | 36 | 65
  SARS-Cov-2 D614G at Month 4-Total: number analyzed (Participants) | 18 | 43 | 50 | 116
  SARS-Cov-2 D614G at Month 4-Total | 17 | 36 | 46 | 108
  SARS-Cov-2 D614G at Month 4-non-RSA: number analyzed (Participants) | 2 | 12 | 13 | 44
  SARS-Cov-2 D614G at Month 4-non-RSA | 2 | 9 | 10 | 43

40. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Days Since SARS-CoV-2 Diagnosis Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and days since SARS-CoV-2 diagnosis group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 49 | 83 | 76 | 161
Titer
  SARS-Cov-2 D614G-ID50 at Month 0-RSA: number analyzed (Participants) | 22 | 51 | 54 | 109
  SARS-Cov-2 D614G-ID50 at Month 0-RSA | 341.2 [110.2 to 1948.9] | 312.2 [149.5 to 1607.4] | 269.1 [127.5 to 884.9] | 320.3 [115.3 to 1045.8]
  SARS-Cov-2 D614G-ID50 at Month 0-Total: number analyzed (Participants) | 24 | 68 | 71 | 157
  SARS-Cov-2 D614G-ID50 at Month 0-Total | 341.2 [80.9 to 1945.6] | 296.6 [116.6 to 1463.5] | 240.7 [74.5 to 903] | 360.1 [93.9 to 1149]
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA: number analyzed (Participants) | 2 | 17 | 17 | 48
  SARS-Cov-2 D614G-ID50 at Month 0-non-RSA | 252.2 [158.5 to 345.9] | 220.2 [10 to 329.4] | 57.2 [5 to 909.9] | 416.1 [82.3 to 1386.4]
  SARS-Cov-2 D614G-ID50 at Month 12-RSA: number analyzed (Participants) | 7 | 22 | 24 | 58
  SARS-Cov-2 D614G-ID50 at Month 12-RSA | 7856.6 [3305.9 to 16483.5] | 1884.6 [512 to 11721.5] | 1657.3 [346.8 to 6270.6] | 1591.4 [256.7 to 9041.5]
  SARS-Cov-2 D614G-ID50 at Month 12-Total: number analyzed (Participants) | 9 | 34 | 38 | 99
  SARS-Cov-2 D614G-ID50 at Month 12-Total | 6035.4 [576.3 to 9886.8] | 1436.1 [297.4 to 6307.1] | 600.3 [233.6 to 3294.7] | 1194.2 [285.7 to 7388.6]
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA: number analyzed (Participants) | 2 | 12 | 14 | 41
  SARS-Cov-2 D614G-ID50 at Month 12-non-RSA | 964.7 [487.3 to 1442] | 347.6 [275.1 to 1767.6] | 408.4 [218.3 to 1370.6] | 872 [358 to 6952.5]
  SARS-Cov-2 D614G-ID50 at Month 2-RSA: number analyzed (Participants) | 16 | 31 | 40 | 70
  SARS-Cov-2 D614G-ID50 at Month 2-RSA | 244.3 [55.8 to 554.9] | 147.5 [60.9 to 878.4] | 156.1 [67.4 to 472.6] | 223.1 [58.9 to 584.3]
  SARS-Cov-2 D614G-ID50 at Month 2-Total: number analyzed (Participants) | 18 | 44 | 56 | 118
  SARS-Cov-2 D614G-ID50 at Month 2-Total | 201.6 [52.4 to 494.3] | 98.8 [34.7 to 310.9] | 133.4 [39.3 to 429.7] | 157.5 [54.3 to 477.8]
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA: number analyzed (Participants) | 2 | 13 | 16 | 48
  SARS-Cov-2 D614G-ID50 at Month 2-non-RSA | 100.9 [53 to 148.9] | 36 [5 to 52.4] | 26.4 [7.4 to 263.5] | 124 [48.1 to 360.6]
  SARS-Cov-2 D614G-ID50 at Month 4-RSA: number analyzed (Participants) | 16 | 31 | 37 | 72
  SARS-Cov-2 D614G-ID50 at Month 4-RSA | 279.6 [25.1 to 801.6] | 570.1 [54.3 to 1747.8] | 335.1 [78.9 to 908.3] | 275.6 [90.3 to 706.4]
  SARS-Cov-2 D614G-ID50 at Month 4-Total: number analyzed (Participants) | 18 | 43 | 50 | 116
  SARS-Cov-2 D614G-ID50 at Month 4-Total | 222 [15 to 687.1] | 203.6 [54.3 to 1457.4] | 324.7 [82.6 to 944.1] | 262.9 [84.1 to 705.8]
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA: number analyzed (Participants) | 2 | 12 | 13 | 44
  SARS-Cov-2 D614G-ID50 at Month 4-non-RSA | 86.5 [48.3 to 124.8] | 137.7 [58.8 to 200.4] | 312.5 [208.9 to 1661.1] | 205.5 [69.5 to 563.2]
  SARS-Cov-2 D614G-ID80 at Month 0-RSA: number analyzed (Participants) | 22 | 51 | 54 | 109
  SARS-Cov-2 D614G-ID80 at Month 0-RSA | 100.3 [37.6 to 619.6] | 117.8 [34.6 to 475.7] | 68.2 [34.7 to 201.9] | 77.2 [32.9 to 233.5]
  SARS-Cov-2 D614G-ID80 at Month 0-Total: number analyzed (Participants) | 24 | 68 | 71 | 157
  SARS-Cov-2 D614G-ID80 at Month 0-Total | 98.7 [32.9 to 546.7] | 78.8 [33.4 to 330.7] | 60.3 [27.3 to 196.2] | 81.4 [28.4 to 274.7]
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA: number analyzed (Participants) | 2 | 17 | 17 | 48
  SARS-Cov-2 D614G-ID80 at Month 0-non-RSA | 63.8 [47.9 to 79.8] | 39.7 [10 to 130.8] | 24.5 [5 to 179] | 106.2 [27.5 to 361.3]
  SARS-Cov-2 D614G-ID80 at Month 12-RSA: number analyzed (Participants) | 7 | 22 | 24 | 58
  SARS-Cov-2 D614G-ID80 at Month 12-RSA | 2749.2 [590.8 to 4116.1] | 495.1 [178.3 to 1335.7] | 410.6 [115.5 to 1749.9] | 351.6 [60.4 to 2756.9]
  SARS-Cov-2 D614G-ID80 at Month 12-Total: number analyzed (Participants) | 9 | 34 | 38 | 99
  SARS-Cov-2 D614G-ID80 at Month 12-Total | 1076.7 [104.9 to 2760.8] | 390.9 [114.7 to 1196.3] | 182.2 [62.2 to 794.2] | 250.7 [83.5 to 2250.8]
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA: number analyzed (Participants) | 2 | 12 | 14 | 41
  SARS-Cov-2 D614G-ID80 at Month 12-non-RSA | 361.3 [185.7 to 537] | 133.8 [101.6 to 605.3] | 119.1 [62.2 to 346] | 238.8 [103.1 to 1837]
  SARS-Cov-2 D614G-ID80 at Month 2-RSA: number analyzed (Participants) | 16 | 31 | 40 | 70
  SARS-Cov-2 D614G-ID80 at Month 2-RSA | 55.8 [10 to 131.9] | 39.3 [14.4 to 197.3] | 36.6 [12.5 to 116.9] | 60.4 [23.4 to 158.4]
  SARS-Cov-2 D614G-ID80 at Month 2-Total: number analyzed (Participants) | 18 | 44 | 56 | 118
  SARS-Cov-2 D614G-ID80 at Month 2-Total | 40.1 [10 to 114.1] | 34.7 [10 to 83.7] | 34.9 [10 to 93] | 41.2 [10.7 to 140]
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA: number analyzed (Participants) | 2 | 13 | 16 | 48
  SARS-Cov-2 D614G-ID80 at Month 2-non-RSA | 19.8 [12.4 to 27.3] | 10 [5 to 24.5] | 16.2 [6.9 to 54.6] | 32.3 [10 to 112.7]
  SARS-Cov-2 D614G-ID80 at Month 4-RSA: number analyzed (Participants) | 16 | 31 | 37 | 72
  SARS-Cov-2 D614G-ID80 at Month 4-RSA | 71.4 [10 to 150.1] | 147.2 [15.9 to 398.2] | 120.5 [30.9 to 215.9] | 86.5 [32.4 to 180.7]
  SARS-Cov-2 D614G-ID80 at Month 4-Total: number analyzed (Participants) | 18 | 43 | 50 | 116
  SARS-Cov-2 D614G-ID80 at Month 4-Total | 54 [10 to 134.1] | 54.1 [15.9 to 339.6] | 119.9 [31.1 to 232] | 73.7 [26.7 to 180.7]
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA: number analyzed (Participants) | 2 | 12 | 13 | 44
  SARS-Cov-2 D614G-ID80 at Month 4-non-RSA | 23.3 [16.6 to 29.9] | 40 [21.2 to 47] | 119.2 [43.3 to 363.7] | 50.5 [24.2 to 180]

41. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (ADCC) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by antibody-dependent cellular cytotoxicity assay (ADCC) at Visit 1, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort (USA and Peru)
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 24 | 58 | 64 | 110
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 12 | 38 | 33 | 69
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 24 | 58 | 64 | 110
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 16 | 39 | 38 | 60

42. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (ADCC) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by antibody-dependent cellular cytotoxicity assay (ADCC) Visit 1, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: Percent CD107a+ NK Cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Percent CD107a+ NK Cells
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total: number analyzed (Participants) | 24 | 58 | 64 | 110
  Bkg. Subtracted CD107A NK Cells-I-ADCC at Month 0-Total | 4.1 [0.9 to 6.4] | 7.2 [1.5 to 14.6] | 5.6 [1.1 to 13.3] | 6.3 [2.2 to 14.6]
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total: number analyzed (Participants) | 24 | 58 | 64 | 110
  Bkg. Subtracted CD107A NK Cells-T-ADCC at Month 0-Total | 6.5 [4.7 to 13.7] | 9.7 [3.7 to 15.3] | 6.9 [2.9 to 14.1] | 5.8 [2.8 to 11.3]

43. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate (ICS) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate by flow cytometry at Visit 1, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0
Population: American Population with positive responders (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
Participants
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD4+-Any COV2 at Month 0-Peru | 17 | 40 | 41 | 45
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 30 | 80 | 88 | 167
  CD4+-Any COV2 at Month 0-Total | 22 | 58 | 66 | 126
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 36 | 113
  CD4+-Any COV2 at Month 0-USA | 5 | 18 | 25 | 81
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 21 | 47 | 52 | 54
  CD4+-E M at Month 0-Peru | 10 | 37 | 32 | 36
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 29 | 78 | 88 | 163
  CD4+-E M at Month 0-Total | 12 | 50 | 47 | 94
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 8 | 31 | 36 | 109
  CD4+-E M at Month 0-USA | 2 | 13 | 15 | 58
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD4+-N at Month 0-Peru | 14 | 37 | 30 | 35
  CD4+-N at Month 0-Total: number analyzed (Participants) | 29 | 80 | 88 | 167
  CD4+-N at Month 0-Total | 16 | 49 | 51 | 105
  CD4+-N at Month 0-USA: number analyzed (Participants) | 8 | 31 | 36 | 113
  CD4+-N at Month 0-USA | 2 | 12 | 21 | 70
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 51 | 52
  CD4+-ORF3a6 at Month 0-Peru | 4 | 21 | 22 | 18
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 29 | 79 | 87 | 162
  CD4+-ORF3a6 at Month 0-Total | 5 | 26 | 32 | 63
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 8 | 31 | 36 | 110
  CD4+-ORF3a6 at Month 0-USA | 1 | 5 | 10 | 45
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 52 | 53
  CD4+-ORF7a7b8 at Month 0-Peru | 8 | 29 | 26 | 23
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 28 | 79 | 88 | 161
  CD4+-ORF7a7b8 at Month 0-Total | 9 | 34 | 35 | 64
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 7 | 31 | 36 | 108
  CD4+-ORF7a7b8 at Month 0-USA | 1 | 5 | 9 | 41
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 51 | 53
  CD4+-S1 at Month 0-Peru | 12 | 39 | 34 | 41
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 30 | 79 | 87 | 165
  CD4+-S1 at Month 0-Total | 16 | 53 | 53 | 109
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 36 | 112
  CD4+-S1 at Month 0-USA | 4 | 14 | 19 | 68
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD4+-S2 at Month 0-Peru | 13 | 37 | 34 | 32
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 30 | 80 | 88 | 167
  CD4+-S2 at Month 0-Total | 17 | 48 | 54 | 100
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 9 | 31 | 36 | 113
  CD4+-S2 at Month 0-USA | 4 | 11 | 20 | 68
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD4+-Spike at Month 0-Peru | 15 | 40 | 38 | 42
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 30 | 80 | 88 | 167
  CD4+-Spike at Month 0-Total | 20 | 54 | 61 | 117
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 9 | 31 | 36 | 113
  CD4+-Spike at Month 0-USA | 5 | 14 | 23 | 75
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD8+-Any COV2 at Month 0-Peru | 12 | 34 | 42 | 34
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 30 | 79 | 88 | 167
  CD8+-Any COV2 at Month 0-Total | 17 | 53 | 64 | 98
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 9 | 30 | 36 | 113
  CD8+-Any COV2 at Month 0-USA | 5 | 19 | 22 | 64
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 52 | 54
  CD8+-E M at Month 0-Peru | 0 | 3 | 7 | 3
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 29 | 78 | 88 | 163
  CD8+-E M at Month 0-Total | 1 | 4 | 8 | 17
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 8 | 30 | 36 | 109
  CD8+-E M at Month 0-USA | 1 | 1 | 1 | 14
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD8+-N at Month 0-Peru | 11 | 31 | 41 | 25
  CD8+-N at Month 0-Total: number analyzed (Participants) | 29 | 79 | 88 | 167
  CD8+-N at Month 0-Total | 16 | 45 | 61 | 78
  CD8+-N at Month 0-USA: number analyzed (Participants) | 8 | 30 | 36 | 113
  CD8+-N at Month 0-USA | 5 | 14 | 20 | 53
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 52 | 53
  CD8+-ORF3a6 at Month 0-Peru | 4 | 9 | 23 | 14
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 29 | 78 | 88 | 163
  CD8+-ORF3a6 at Month 0-Total | 5 | 13 | 30 | 32
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 8 | 30 | 36 | 110
  CD8+-ORF3a6 at Month 0-USA | 1 | 4 | 7 | 18
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 52 | 53
  CD8+-ORF7a7b8 at Month 0-Peru | 2 | 12 | 23 | 14
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 28 | 78 | 88 | 160
  CD8+-ORF7a7b8 at Month 0-Total | 2 | 16 | 25 | 28
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 7 | 30 | 36 | 107
  CD8+-ORF7a7b8 at Month 0-USA | 0 | 4 | 2 | 14
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 21 | 48 | 51 | 54
  CD8+-S1 at Month 0-Peru | 2 | 15 | 11 | 14
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 30 | 78 | 87 | 166
  CD8+-S1 at Month 0-Total | 2 | 20 | 17 | 32
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 9 | 30 | 36 | 112
  CD8+-S1 at Month 0-USA | 0 | 5 | 6 | 18
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 51 | 54
  CD8+-S2 at Month 0-Peru | 2 | 8 | 2 | 6
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 30 | 79 | 87 | 167
  CD8+-S2 at Month 0-Total | 2 | 11 | 2 | 15
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 9 | 30 | 36 | 113
  CD8+-S2 at Month 0-USA | 0 | 3 | 0 | 9
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 21 | 49 | 52 | 54
  CD8+-Spike at Month 0-Peru | 3 | 16 | 12 | 16
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 30 | 79 | 88 | 167
  CD8+-Spike at Month 0-Total | 3 | 23 | 18 | 38
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 9 | 30 | 36 | 113
  CD8+-Spike at Month 0-USA | 0 | 7 | 6 | 22

44. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude (ICS) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and days since SARS-CoV-2 diagnosis group among America Cohort
Time Frame: Measured at Months 0
Population: American Population with positive responders (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: % T cells expressing IFN-g/IL-2
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
% T cells expressing IFN-g/IL-2
  CD4+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 17 | 40 | 41 | 45
  CD4+-Any COV2 at Month 0-Peru | 0.4 [0.2 to 0.7] | 1 [0.6 to 1.6] | 0.8 [0.3 to 1.3] | 0.6 [0.4 to 1]
  CD4+-Any COV2 at Month 0-Total: number analyzed (Participants) | 22 | 58 | 66 | 126
  CD4+-Any COV2 at Month 0-Total | 0.4 [0.2 to 0.7] | 0.8 [0.4 to 1.5] | 0.6 [0.2 to 1.1] | 0.6 [0.4 to 1]
  CD4+-Any COV2 at Month 0-USA: number analyzed (Participants) | 5 | 18 | 25 | 81
  CD4+-Any COV2 at Month 0-USA | 0.3 [0.2 to 0.6] | 0.3 [0.3 to 0.7] | 0.4 [0.2 to 0.8] | 0.6 [0.4 to 1]
  CD4+-E M at Month 0-Peru: number analyzed (Participants) | 10 | 37 | 32 | 36
  CD4+-E M at Month 0-Peru | 0.1 [0.1 to 0.3] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M at Month 0-Total: number analyzed (Participants) | 12 | 50 | 47 | 94
  CD4+-E M at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2]
  CD4+-E M at Month 0-USA: number analyzed (Participants) | 2 | 13 | 15 | 58
  CD4+-E M at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  CD4+-N at Month 0-Peru: number analyzed (Participants) | 14 | 37 | 30 | 35
  CD4+-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-Total: number analyzed (Participants) | 16 | 49 | 51 | 105
  CD4+-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N at Month 0-USA: number analyzed (Participants) | 2 | 12 | 21 | 70
  CD4+-N at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 4 | 21 | 22 | 18
  CD4+-ORF3a6 at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 5 | 26 | 32 | 63
  CD4+-ORF3a6 at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 1 | 5 | 10 | 45
  CD4+-ORF3a6 at Month 0-USA | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 8 | 29 | 26 | 23
  CD4+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 9 | 34 | 35 | 64
  CD4+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 1 | 5 | 9 | 41
  CD4+-ORF7a7b8 at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  CD4+-S1 at Month 0-Peru: number analyzed (Participants) | 12 | 39 | 34 | 41
  CD4+-S1 at Month 0-Peru | 0.2 [0.1 to 0.2] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3]
  CD4+-S1 at Month 0-Total: number analyzed (Participants) | 16 | 53 | 53 | 109
  CD4+-S1 at Month 0-Total | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3]
  CD4+-S1 at Month 0-USA: number analyzed (Participants) | 4 | 14 | 19 | 68
  CD4+-S1 at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD4+-S2 at Month 0-Peru: number analyzed (Participants) | 13 | 37 | 34 | 32
  CD4+-S2 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2 at Month 0-Total: number analyzed (Participants) | 17 | 48 | 54 | 100
  CD4+-S2 at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2 at Month 0-USA: number analyzed (Participants) | 4 | 11 | 20 | 68
  CD4+-S2 at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-Spike at Month 0-Peru: number analyzed (Participants) | 15 | 40 | 38 | 42
  CD4+-Spike at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.4 [0.3 to 0.7] | 0.4 [0.2 to 0.7] | 0.3 [0.2 to 0.5]
  CD4+-Spike at Month 0-Total: number analyzed (Participants) | 20 | 54 | 61 | 117
  CD4+-Spike at Month 0-Total | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.6] | 0.3 [0.1 to 0.5] | 0.3 [0.2 to 0.5]
  CD4+-Spike at Month 0-USA: number analyzed (Participants) | 5 | 14 | 23 | 75
  CD4+-Spike at Month 0-USA | 0.1 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.5]
  CD8+-Any COV2 at Month 0-Peru: number analyzed (Participants) | 12 | 34 | 42 | 34
  CD8+-Any COV2 at Month 0-Peru | 0.3 [0.2 to 0.4] | 0.5 [0.3 to 1.4] | 0.7 [0.4 to 1.6] | 0.4 [0.2 to 1.2]
  CD8+-Any COV2 at Month 0-Total: number analyzed (Participants) | 17 | 53 | 64 | 98
  CD8+-Any COV2 at Month 0-Total | 0.2 [0.2 to 0.3] | 0.4 [0.2 to 0.8] | 0.5 [0.3 to 1.1] | 0.4 [0.2 to 0.9]
  CD8+-Any COV2 at Month 0-USA: number analyzed (Participants) | 5 | 19 | 22 | 64
  CD8+-Any COV2 at Month 0-USA | 0.2 [0.2 to 0.2] | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.3] | 0.4 [0.2 to 0.8]
  CD8+-E M at Month 0-Peru: number analyzed (Participants) | 0 | 3 | 7 | 3
  CD8+-E M at Month 0-Peru |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.3 [0.2 to 0.4]
  CD8+-E M at Month 0-Total: number analyzed (Participants) | 1 | 4 | 8 | 17
  CD8+-E M at Month 0-Total | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.3]
  CD8+-E M at Month 0-USA: number analyzed (Participants) | 1 | 1 | 1 | 14
  CD8+-E M at Month 0-USA | 0.2 [0.2 to 0.2] | 0 [0 to 0] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD8+-N at Month 0-Peru: number analyzed (Participants) | 11 | 31 | 41 | 25
  CD8+-N at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.4 [0.2 to 1] | 0.3 [0.1 to 0.9]
  CD8+-N at Month 0-Total: number analyzed (Participants) | 16 | 45 | 61 | 78
  CD8+-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6]
  CD8+-N at Month 0-USA: number analyzed (Participants) | 5 | 14 | 20 | 53
  CD8+-N at Month 0-USA | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4]
  CD8+-ORF3a6 at Month 0-Peru: number analyzed (Participants) | 4 | 9 | 23 | 14
  CD8+-ORF3a6 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.2 to 0.6] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.6]
  CD8+-ORF3a6 at Month 0-Total: number analyzed (Participants) | 5 | 13 | 30 | 32
  CD8+-ORF3a6 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5]
  CD8+-ORF3a6 at Month 0-USA: number analyzed (Participants) | 1 | 4 | 7 | 18
  CD8+-ORF3a6 at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.3 [0.2 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+-ORF7a7b8 at Month 0-Peru: number analyzed (Participants) | 2 | 12 | 23 | 14
  CD8+-ORF7a7b8 at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.8] | 0.2 [0.1 to 0.7]
  CD8+-ORF7a7b8 at Month 0-Total: number analyzed (Participants) | 2 | 16 | 25 | 28
  CD8+-ORF7a7b8 at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.3] | 0.3 [0.2 to 0.8] | 0.2 [0.1 to 0.6]
  CD8+-ORF7a7b8 at Month 0-USA: number analyzed (Participants) | 0 | 4 | 2 | 14
  CD8+-ORF7a7b8 at Month 0-USA |  | 0.1 [0.1 to 0.1] | 0.6 [0.5 to 0.6] | 0.1 [0.1 to 0.5]
  CD8+-S1 at Month 0-Peru: number analyzed (Participants) | 2 | 15 | 11 | 14
  CD8+-S1 at Month 0-Peru | 0.5 [0.3 to 0.7] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD8+-S1 at Month 0-Total: number analyzed (Participants) | 2 | 20 | 17 | 32
  CD8+-S1 at Month 0-Total | 0.5 [0.3 to 0.7] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S1 at Month 0-USA: number analyzed (Participants) | 0 | 5 | 6 | 18
  CD8+-S1 at Month 0-USA |  | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.3]
  CD8+-S2 at Month 0-Peru: number analyzed (Participants) | 2 | 8 | 2 | 6
  CD8+-S2 at Month 0-Peru | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD8+-S2 at Month 0-Total: number analyzed (Participants) | 2 | 11 | 2 | 15
  CD8+-S2 at Month 0-Total | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.5] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD8+-S2 at Month 0-USA: number analyzed (Participants) | 0 | 3 | 0 | 9
  CD8+-S2 at Month 0-USA |  | 0.2 [0.1 to 0.5] |  | 0.1 [0.1 to 0.1]
  CD8+-Spike at Month 0-Peru: number analyzed (Participants) | 3 | 16 | 12 | 16
  CD8+-Spike at Month 0-Peru | 0.1 [0.1 to 0.7] | 0.3 [0.2 to 0.6] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD8+-Spike at Month 0-Total: number analyzed (Participants) | 3 | 23 | 18 | 38
  CD8+-Spike at Month 0-Total | 0.1 [0.1 to 0.7] | 0.2 [0.1 to 0.5] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-Spike at Month 0-USA: number analyzed (Participants) | 0 | 7 | 6 | 22
  CD8+-Spike at Month 0-USA |  | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3]

45. Primary Outcome: SARS-CoV-2-specific Memory B Cell Response Magnitude (B Cell) by Region and Days Since SARS-CoV-2 Diagnosis Group Among America Cohort
Description: SARS-CoV-2-specific B cell responses and B cell phenotypic data was identified and characterized using fluorescently-labelled recombinant Env proteins (S6P and RBD) in combination with a flow cytometry antibody panel on all available samples from the enrollment visit (V1). The sample will be included in the analysis only if the number of IgD- B cells is equal or greater than 1000 for that sample.
  The table summarized SARS-CoV-2-specific Memory B Cell Response Magnitude (B Cell) by Region and Days Since SARS-CoV-2 Diagnosis Group among America Cohort
Time Frame: Measured at Months 0
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 37 | 88 | 92 | 171
percentage of cells
  %RBD+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %RBD+ IgA+ of Memory B Cells-Peru | 0.01 [0 to 0.03] | 0.01 [0 to 0.06] | 0.01 [0 to 0.03] | 0.02 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %RBD+ IgA+ of Memory B Cells-Total | 0.01 [0 to 0.03] | 0.01 [0 to 0.07] | 0.01 [0 to 0.03] | 0 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %RBD+ IgA+ of Memory B Cells-USA | 0.02 [0.01 to 0.03] | 0.02 [0 to 0.07] | 0.01 [0 to 0.04] | 0 [0 to 0.02]
  %RBD+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %RBD+ IgG+ of Memory B Cells-Peru | 0.1 [0.05 to 0.16] | 0.15 [0.08 to 0.31] | 0.13 [0.06 to 0.29] | 0.29 [0.14 to 0.37]
  %RBD+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %RBD+ IgG+ of Memory B Cells-Total | 0.14 [0.06 to 0.21] | 0.13 [0.06 to 0.27] | 0.13 [0.05 to 0.28] | 0.2 [0.06 to 0.36]
  %RBD+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %RBD+ IgG+ of Memory B Cells-USA | 0.22 [0.13 to 0.31] | 0.12 [0.05 to 0.2] | 0.14 [0.04 to 0.24] | 0.16 [0.04 to 0.33]
  %RBD+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %RBD+ IgM+ of Memory B Cells-Peru | 0 [0 to 0.01] | 0.01 [0 to 0.03] | 0 [0 to 0.01] | 0 [0 to 0]
  %RBD+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %RBD+ IgM+ of Memory B Cells-Total | 0 [0 to 0.01] | 0.01 [0 to 0.03] | 0 [0 to 0.01] | 0 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %RBD+ IgM+ of Memory B Cells-USA | 0.01 [0 to 0.02] | 0.01 [0 to 0.05] | 0 [0 to 0.02] | 0 [0 to 0.01]
  %RBD+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %RBD+ of Total B Cells-Peru | 0.05 [0.03 to 0.07] | 0.08 [0.05 to 0.16] | 0.07 [0.04 to 0.11] | 0.11 [0.07 to 0.16]
  %RBD+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %RBD+ of Total B Cells-Total | 0.06 [0.04 to 0.08] | 0.07 [0.04 to 0.16] | 0.06 [0.03 to 0.11] | 0.07 [0.03 to 0.12]
  %RBD+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %RBD+ of Total B Cells-USA | 0.07 [0.06 to 0.12] | 0.05 [0.04 to 0.17] | 0.04 [0.02 to 0.08] | 0.05 [0.03 to 0.09]
  %S+ IgA+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgA+ of Memory B Cells-Peru | 0.09 [0.05 to 0.14] | 0.08 [0.03 to 0.12] | 0.07 [0.03 to 0.12] | 0.06 [0.03 to 0.12]
  %S+ IgA+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgA+ of Memory B Cells-Total | 0.08 [0.04 to 0.13] | 0.08 [0.03 to 0.13] | 0.06 [0.03 to 0.11] | 0.06 [0.02 to 0.1]
  %S+ IgA+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgA+ of Memory B Cells-USA | 0.05 [0.04 to 0.08] | 0.08 [0.03 to 0.14] | 0.05 [0.02 to 0.09] | 0.06 [0.02 to 0.1]
  %S+ IgA+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgA+ of Total B Cells-Peru | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.01 [0.01 to 0.03]
  %S+ IgA+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgA+ of Total B Cells-Total | 0.02 [0.01 to 0.02] | 0.01 [0.01 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.02]
  %S+ IgA+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgA+ of Total B Cells-USA | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02]
  %S+ IgG+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgG+ of Memory B Cells-Peru | 0.48 [0.33 to 0.95] | 0.77 [0.4 to 1.22] | 0.62 [0.33 to 1.15] | 1 [0.62 to 1.4]
  %S+ IgG+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgG+ of Memory B Cells-Total | 0.52 [0.32 to 1.03] | 0.5 [0.31 to 1] | 0.62 [0.32 to 1.07] | 0.95 [0.38 to 1.44]
  %S+ IgG+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgG+ of Memory B Cells-USA | 0.77 [0.29 to 1.13] | 0.34 [0.13 to 0.56] | 0.6 [0.29 to 0.97] | 0.86 [0.31 to 1.47]
  %S+ IgG+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgG+ of Total B Cells-Peru | 0.11 [0.06 to 0.25] | 0.18 [0.08 to 0.26] | 0.17 [0.11 to 0.29] | 0.21 [0.12 to 0.29]
  %S+ IgG+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgG+ of Total B Cells-Total | 0.13 [0.06 to 0.23] | 0.11 [0.06 to 0.21] | 0.15 [0.06 to 0.25] | 0.16 [0.07 to 0.24]
  %S+ IgG+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgG+ of Total B Cells-USA | 0.15 [0.1 to 0.17] | 0.07 [0.01 to 0.11] | 0.08 [0.04 to 0.11] | 0.13 [0.06 to 0.22]
  %S+ IgM+ IgD+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgM+ IgD+ of Total B Cells-Peru | 0.13 [0.1 to 0.15] | 0.13 [0.09 to 0.16] | 0.1 [0.07 to 0.14] | 0.11 [0.08 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgM+ IgD+ of Total B Cells-Total | 0.11 [0.06 to 0.13] | 0.11 [0.08 to 0.16] | 0.09 [0.07 to 0.13] | 0.1 [0.07 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgM+ IgD+ of Total B Cells-USA | 0.09 [0.06 to 0.1] | 0.1 [0.08 to 0.12] | 0.09 [0.06 to 0.11] | 0.09 [0.07 to 0.14]
  %S+ IgM+ of Memory B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgM+ of Memory B Cells-Peru | 0.06 [0.03 to 0.14] | 0.06 [0.03 to 0.11] | 0.04 [0.01 to 0.06] | 0.02 [0 to 0.04]
  %S+ IgM+ of Memory B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgM+ of Memory B Cells-Total | 0.05 [0.02 to 0.12] | 0.06 [0.03 to 0.11] | 0.04 [0.02 to 0.06] | 0.03 [0 to 0.06]
  %S+ IgM+ of Memory B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgM+ of Memory B Cells-USA | 0.05 [0.02 to 0.08] | 0.06 [0.04 to 0.12] | 0.05 [0.02 to 0.08] | 0.03 [0 to 0.07]
  %S+ IgM+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ IgM+ of Total B Cells-Peru | 0.01 [0 to 0.03] | 0.01 [0.01 to 0.03] | 0.01 [0 to 0.02] | 0 [0 to 0.01]
  %S+ IgM+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ IgM+ of Total B Cells-Total | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0 [0 to 0.01]
  %S+ IgM+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ IgM+ of Total B Cells-USA | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0 [0 to 0.01]
  %S+ of Total B Cells-Peru: number analyzed (Participants) | 18 | 43 | 44 | 41
  %S+ of Total B Cells-Peru | 0.33 [0.2 to 0.51] | 0.43 [0.28 to 0.56] | 0.4 [0.28 to 0.52] | 0.42 [0.3 to 0.52]
  %S+ of Total B Cells-Total: number analyzed (Participants) | 26 | 68 | 70 | 127
  %S+ of Total B Cells-Total | 0.32 [0.22 to 0.42] | 0.32 [0.21 to 0.51] | 0.32 [0.21 to 0.48] | 0.33 [0.21 to 0.5]
  %S+ of Total B Cells-USA: number analyzed (Participants) | 8 | 25 | 26 | 86
  %S+ of Total B Cells-USA | 0.32 [0.28 to 0.34] | 0.24 [0.15 to 0.36] | 0.25 [0.17 to 0.28] | 0.3 [0.2 to 0.48]

46. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG1) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3 , overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2, 4
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Cigarette smoking - current
- Group 2: Cigarette smoking - ever
- Group 3: Marijuana smoking - current
- Group 4: Marijuana smoking - ever
- Group 5: Smoking - any history
- Group 6: Any targeted conditions at enrollment
- Group 7: COPD/emphysema/ asthma
- Group 8: Diabetes
- Group 9: HIV
- Group 10: Hypertension
- Group 11: Immune system disorders
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
Participants
  2019-nCoV S/293F-50-N at Month 0-Peru: number analyzed (Participants) | 148 | 106 | 152 | 146 | 105 | 96 | 144 | 137 | 137 | 131 | 129
  2019-nCoV S/293F-50-N at Month 0-Peru | 143 | 104 | 147 | 141 | 103 | 95 | 140 | 132 | 132 | 129 | 124
  2019-nCoV S/293F-50-N at Month 0-Total: number analyzed (Participants) | 264 | 190 | 268 | 218 | 162 | 139 | 256 | 245 | 241 | 217 | 219
  2019-nCoV S/293F-50-N at Month 0-Total | 248 | 181 | 252 | 206 | 157 | 136 | 241 | 228 | 224 | 210 | 204
  2019-nCoV S/293F-50-N at Month 0-USA: number analyzed (Participants) | 116 | 84 | 116 | 72 | 57 | 43 | 112 | 108 | 104 | 86 | 90
  2019-nCoV S/293F-50-N at Month 0-USA | 105 | 77 | 105 | 65 | 54 | 41 | 101 | 96 | 92 | 81 | 80
  2019-nCoV S/293F-50-N at Month 2-Peru: number analyzed (Participants) | 133 | 96 | 139 | 131 | 95 | 87 | 132 | 124 | 129 | 118 | 121
  2019-nCoV S/293F-50-N at Month 2-Peru | 126 | 93 | 132 | 125 | 92 | 84 | 126 | 117 | 122 | 114 | 114
  2019-nCoV S/293F-50-N at Month 2-Total: number analyzed (Participants) | 253 | 179 | 261 | 200 | 148 | 131 | 243 | 237 | 245 | 201 | 220
  2019-nCoV S/293F-50-N at Month 2-Total | 235 | 168 | 241 | 187 | 141 | 124 | 224 | 216 | 224 | 190 | 201
  2019-nCoV S/293F-50-N at Month 2-USA: number analyzed (Participants) | 120 | 83 | 122 | 69 | 53 | 44 | 111 | 113 | 116 | 83 | 99
  2019-nCoV S/293F-50-N at Month 2-USA | 109 | 75 | 109 | 62 | 49 | 40 | 98 | 99 | 102 | 76 | 87
  2019-nCoV S/293F-50-N at Month 4-Peru: number analyzed (Participants) | 110 | 83 | 115 | 108 | 82 | 75 | 109 | 103 | 109 | 96 | 104
  2019-nCoV S/293F-50-N at Month 4-Peru | 102 | 79 | 107 | 101 | 78 | 72 | 102 | 95 | 101 | 92 | 96
  2019-nCoV S/293F-50-N at Month 4-Total: number analyzed (Participants) | 189 | 139 | 192 | 158 | 123 | 103 | 182 | 178 | 183 | 146 | 169
  2019-nCoV S/293F-50-N at Month 4-Total | 172 | 130 | 173 | 145 | 116 | 98 | 164 | 160 | 164 | 139 | 151
  2019-nCoV S/293F-50-N at Month 4-USA: number analyzed (Participants) | 79 | 56 | 77 | 50 | 41 | 28 | 73 | 75 | 74 | 50 | 65
  2019-nCoV S/293F-50-N at Month 4-USA | 70 | 51 | 66 | 44 | 38 | 26 | 62 | 65 | 63 | 47 | 55
  2019-nCoV S/293F-50-Y at Month 0-Peru: number analyzed (Participants) | 4 | 46 | 0 | 6 | 47 | 56 | 8 | 15 | 15 | 21 | 23
  2019-nCoV S/293F-50-Y at Month 0-Peru | 4 | 43 | 0 | 6 | 44 | 52 | 7 | 15 | 15 | 18 | 23
  2019-nCoV S/293F-50-Y at Month 0-Total: number analyzed (Participants) | 20 | 94 | 16 | 66 | 122 | 145 | 28 | 39 | 43 | 67 | 65
  2019-nCoV S/293F-50-Y at Month 0-Total | 16 | 83 | 12 | 58 | 107 | 128 | 23 | 36 | 40 | 54 | 60
  2019-nCoV S/293F-50-Y at Month 0-USA: number analyzed (Participants) | 16 | 48 | 16 | 60 | 75 | 89 | 20 | 24 | 28 | 46 | 42
  2019-nCoV S/293F-50-Y at Month 0-USA | 12 | 40 | 12 | 52 | 63 | 76 | 16 | 21 | 25 | 36 | 37
  2019-nCoV S/293F-50-Y at Month 2-Peru: number analyzed (Participants) | 6 | 43 | 0 | 8 | 44 | 52 | 7 | 15 | 10 | 21 | 18
  2019-nCoV S/293F-50-Y at Month 2-Peru | 6 | 39 | 0 | 7 | 40 | 48 | 6 | 15 | 10 | 18 | 18
  2019-nCoV S/293F-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 11 | 72 | 124 | 141 | 29 | 35 | 27 | 71 | 52
  2019-nCoV S/293F-50-Y at Month 2-Total | 15 | 82 | 9 | 63 | 109 | 126 | 26 | 34 | 26 | 60 | 49
  2019-nCoV S/293F-50-Y at Month 2-USA: number analyzed (Participants) | 13 | 50 | 11 | 64 | 80 | 89 | 22 | 20 | 17 | 50 | 34
  2019-nCoV S/293F-50-Y at Month 2-USA | 9 | 43 | 9 | 56 | 69 | 78 | 20 | 19 | 16 | 42 | 31
  2019-nCoV S/293F-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 32 | 0 | 7 | 33 | 40 | 6 | 12 | 6 | 19 | 11
  2019-nCoV S/293F-50-Y at Month 4-Peru | 5 | 28 | 0 | 6 | 29 | 35 | 5 | 12 | 6 | 15 | 11
  2019-nCoV S/293F-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 99 | 20 | 24 | 19 | 56 | 33
  2019-nCoV S/293F-50-Y at Month 4-Total | 11 | 53 | 10 | 38 | 67 | 85 | 19 | 23 | 19 | 44 | 32
  2019-nCoV S/293F-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 59 | 14 | 12 | 13 | 37 | 22
  2019-nCoV S/293F-50-Y at Month 4-USA | 6 | 25 | 10 | 32 | 38 | 50 | 14 | 11 | 13 | 29 | 21
  SARS-CoV-2 DB His-50-N at Month 0-Peru: number analyzed (Participants) | 167 | 123 | 174 | 165 | 122 | 113 | 165 | 159 | 159 | 149 | 151
  SARS-CoV-2 DB His-50-N at Month 0-Peru | 156 | 116 | 163 | 155 | 115 | 108 | 155 | 148 | 148 | 143 | 140
  SARS-CoV-2 DB His-50-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 346 | 268 | 204 | 188 | 328 | 324 | 324 | 280 | 293
  SARS-CoV-2 DB His-50-N at Month 0-Total | 306 | 220 | 309 | 241 | 184 | 173 | 291 | 288 | 285 | 259 | 258
  SARS-CoV-2 DB His-50-N at Month 0-USA: number analyzed (Participants) | 176 | 124 | 172 | 103 | 82 | 75 | 163 | 165 | 165 | 131 | 142
  SARS-CoV-2 DB His-50-N at Month 0-USA | 150 | 104 | 146 | 86 | 69 | 65 | 136 | 140 | 137 | 116 | 118
  SARS-CoV-2 DB His-50-N at Month 2-Peru: number analyzed (Participants) | 132 | 97 | 137 | 130 | 96 | 88 | 131 | 122 | 127 | 117 | 120
  SARS-CoV-2 DB His-50-N at Month 2-Peru | 124 | 91 | 129 | 122 | 90 | 83 | 123 | 114 | 119 | 112 | 112
  SARS-CoV-2 DB His-50-N at Month 2-Total: number analyzed (Participants) | 256 | 184 | 261 | 200 | 150 | 136 | 247 | 240 | 248 | 204 | 224
  SARS-CoV-2 DB His-50-N at Month 2-Total | 233 | 166 | 236 | 181 | 136 | 125 | 221 | 214 | 223 | 189 | 201
  SARS-CoV-2 DB His-50-N at Month 2-USA: number analyzed (Participants) | 124 | 87 | 124 | 70 | 54 | 48 | 116 | 118 | 121 | 87 | 104
  SARS-CoV-2 DB His-50-N at Month 2-USA | 109 | 75 | 107 | 59 | 46 | 42 | 98 | 100 | 104 | 77 | 89
  SARS-CoV-2 DB His-50-N at Month 4-Peru: number analyzed (Participants) | 109 | 83 | 114 | 107 | 82 | 75 | 109 | 102 | 108 | 95 | 104
  SARS-CoV-2 DB His-50-N at Month 4-Peru | 100 | 78 | 105 | 99 | 77 | 71 | 101 | 93 | 99 | 90 | 95
  SARS-CoV-2 DB His-50-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 103 | 181 | 177 | 181 | 145 | 168
  SARS-CoV-2 DB His-50-N at Month 4-Total | 167 | 126 | 168 | 140 | 112 | 97 | 159 | 156 | 160 | 136 | 148
  SARS-CoV-2 DB His-50-N at Month 4-USA: number analyzed (Participants) | 78 | 55 | 76 | 49 | 40 | 28 | 72 | 75 | 73 | 50 | 64
  SARS-CoV-2 DB His-50-N at Month 4-USA | 67 | 48 | 63 | 41 | 35 | 26 | 58 | 63 | 61 | 46 | 53
  SARS-CoV-2 DB His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 61 | 9 | 15 | 15 | 25 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Peru | 7 | 47 | 0 | 8 | 48 | 55 | 8 | 15 | 15 | 20 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 21 | 99 | 163 | 179 | 39 | 43 | 43 | 87 | 74
  SARS-CoV-2 DB His-50-Y at Month 0-Total | 20 | 106 | 17 | 85 | 142 | 153 | 35 | 38 | 41 | 67 | 68
  SARS-CoV-2 DB His-50-Y at Month 0-USA: number analyzed (Participants) | 17 | 69 | 21 | 90 | 111 | 118 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 DB His-50-Y at Month 0-USA | 13 | 59 | 17 | 77 | 94 | 98 | 27 | 23 | 26 | 47 | 45
  SARS-CoV-2 DB His-50-Y at Month 2-Peru: number analyzed (Participants) | 5 | 40 | 0 | 7 | 41 | 49 | 6 | 15 | 10 | 20 | 17
  SARS-CoV-2 DB His-50-Y at Month 2-Peru | 5 | 38 | 0 | 7 | 39 | 46 | 6 | 15 | 10 | 17 | 17
  SARS-CoV-2 DB His-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 91 | 14 | 75 | 125 | 139 | 28 | 35 | 27 | 71 | 51
  SARS-CoV-2 DB His-50-Y at Month 2-Total | 14 | 81 | 11 | 66 | 111 | 122 | 26 | 33 | 24 | 58 | 46
  SARS-CoV-2 DB His-50-Y at Month 2-USA: number analyzed (Participants) | 14 | 51 | 14 | 68 | 84 | 90 | 22 | 20 | 17 | 51 | 34
  SARS-CoV-2 DB His-50-Y at Month 2-USA | 9 | 43 | 11 | 59 | 72 | 76 | 20 | 18 | 14 | 41 | 29
  SARS-CoV-2 DB His-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 31 | 0 | 7 | 32 | 39 | 5 | 12 | 6 | 19 | 10
  SARS-CoV-2 DB His-50-Y at Month 4-Peru | 5 | 27 | 0 | 6 | 28 | 34 | 4 | 12 | 6 | 15 | 10
  SARS-CoV-2 DB His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 97 | 19 | 23 | 19 | 55 | 32
  SARS-CoV-2 DB His-50-Y at Month 4-Total | 10 | 51 | 9 | 37 | 65 | 80 | 18 | 21 | 17 | 41 | 29
  SARS-CoV-2 DB His-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 58 | 14 | 11 | 13 | 36 | 22
  SARS-CoV-2 DB His-50-Y at Month 4-USA | 5 | 24 | 9 | 31 | 37 | 46 | 14 | 9 | 11 | 26 | 19
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru: number analyzed (Participants) | 167 | 123 | 174 | 165 | 122 | 113 | 165 | 159 | 159 | 149 | 151
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru | 156 | 116 | 163 | 155 | 115 | 108 | 155 | 148 | 148 | 143 | 140
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 348 | 270 | 205 | 187 | 328 | 323 | 324 | 280 | 293
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total | 306 | 219 | 312 | 244 | 185 | 171 | 290 | 284 | 285 | 257 | 258
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA: number analyzed (Participants) | 176 | 124 | 174 | 105 | 83 | 74 | 163 | 164 | 165 | 131 | 142
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA | 150 | 103 | 149 | 89 | 70 | 63 | 135 | 136 | 137 | 114 | 118
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru: number analyzed (Participants) | 131 | 94 | 136 | 128 | 93 | 87 | 129 | 121 | 127 | 115 | 121
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru | 121 | 88 | 126 | 119 | 87 | 82 | 120 | 111 | 117 | 109 | 111
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total: number analyzed (Participants) | 250 | 176 | 257 | 197 | 146 | 133 | 240 | 235 | 244 | 199 | 222
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total | 225 | 159 | 230 | 179 | 133 | 122 | 213 | 206 | 216 | 182 | 198
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA: number analyzed (Participants) | 119 | 82 | 121 | 69 | 53 | 46 | 111 | 114 | 117 | 84 | 101
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA | 104 | 71 | 104 | 60 | 46 | 40 | 93 | 95 | 99 | 73 | 87
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-Peru: number analyzed (Participants) | 103 | 78 | 108 | 101 | 77 | 72 | 103 | 96 | 102 | 92 | 98
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-Peru | 93 | 72 | 98 | 92 | 71 | 68 | 95 | 86 | 92 | 86 | 88
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-Total: number analyzed (Participants) | 177 | 130 | 180 | 148 | 115 | 98 | 172 | 168 | 172 | 140 | 159
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-Total | 154 | 116 | 155 | 131 | 104 | 91 | 148 | 144 | 147 | 129 | 136
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-USA: number analyzed (Participants) | 74 | 52 | 72 | 47 | 38 | 26 | 69 | 72 | 70 | 48 | 61
  SARS-CoV-2 Nucleoprotein His-50-N at Month 4-USA | 61 | 44 | 57 | 39 | 33 | 23 | 53 | 58 | 55 | 43 | 48
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 61 | 9 | 15 | 15 | 25 | 23
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru | 7 | 47 | 0 | 8 | 48 | 55 | 8 | 15 | 15 | 20 | 23
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 19 | 97 | 162 | 180 | 39 | 44 | 43 | 87 | 74
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total | 18 | 105 | 12 | 80 | 139 | 153 | 34 | 40 | 39 | 67 | 66
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA: number analyzed (Participants) | 17 | 69 | 19 | 88 | 110 | 119 | 30 | 29 | 28 | 62 | 51
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA | 11 | 58 | 12 | 72 | 91 | 98 | 26 | 25 | 24 | 47 | 43
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru: number analyzed (Participants) | 5 | 42 | 0 | 8 | 43 | 49 | 7 | 15 | 9 | 21 | 15
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru | 5 | 38 | 0 | 7 | 39 | 44 | 6 | 15 | 9 | 17 | 15
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 12 | 72 | 123 | 136 | 29 | 34 | 25 | 70 | 47
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total | 14 | 80 | 9 | 60 | 106 | 117 | 26 | 33 | 23 | 57 | 41
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA: number analyzed (Participants) | 14 | 51 | 12 | 64 | 80 | 87 | 22 | 19 | 16 | 49 | 32
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA | 9 | 42 | 9 | 53 | 67 | 73 | 20 | 18 | 14 | 40 | 26
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 30 | 0 | 7 | 31 | 36 | 5 | 12 | 6 | 16 | 10
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-Peru | 5 | 26 | 0 | 6 | 27 | 30 | 3 | 12 | 6 | 12 | 10
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 60 | 10 | 42 | 75 | 92 | 18 | 22 | 18 | 50 | 31
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-Total | 10 | 48 | 9 | 33 | 60 | 73 | 16 | 20 | 17 | 35 | 28
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 30 | 10 | 35 | 44 | 56 | 13 | 10 | 12 | 34 | 21
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 4-USA | 5 | 22 | 9 | 27 | 33 | 43 | 13 | 8 | 11 | 23 | 18
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru: number analyzed (Participants) | 139 | 100 | 140 | 135 | 100 | 86 | 132 | 125 | 125 | 120 | 118
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru | 135 | 98 | 136 | 131 | 98 | 85 | 128 | 121 | 121 | 119 | 114
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total: number analyzed (Participants) | 248 | 180 | 248 | 201 | 154 | 126 | 237 | 226 | 221 | 201 | 200
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total | 232 | 170 | 232 | 188 | 147 | 121 | 221 | 209 | 204 | 193 | 185
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA: number analyzed (Participants) | 109 | 80 | 108 | 66 | 54 | 40 | 105 | 101 | 96 | 81 | 82
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA | 97 | 72 | 96 | 57 | 49 | 36 | 93 | 88 | 83 | 74 | 71
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru: number analyzed (Participants) | 133 | 96 | 138 | 130 | 95 | 87 | 131 | 123 | 128 | 117 | 121
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru | 124 | 90 | 129 | 121 | 89 | 82 | 123 | 114 | 119 | 111 | 112
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total: number analyzed (Participants) | 257 | 183 | 263 | 201 | 150 | 136 | 246 | 240 | 249 | 204 | 225
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total | 236 | 169 | 240 | 185 | 140 | 126 | 223 | 215 | 225 | 190 | 203
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA: number analyzed (Participants) | 124 | 87 | 125 | 71 | 55 | 49 | 115 | 117 | 121 | 87 | 104
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA | 112 | 79 | 111 | 64 | 51 | 44 | 100 | 101 | 106 | 79 | 91
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-Peru: number analyzed (Participants) | 109 | 83 | 114 | 107 | 82 | 74 | 108 | 102 | 108 | 95 | 103
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-Peru | 101 | 79 | 106 | 100 | 78 | 71 | 101 | 94 | 100 | 91 | 95
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 102 | 180 | 177 | 181 | 145 | 167
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-Total | 170 | 129 | 171 | 143 | 115 | 97 | 162 | 159 | 162 | 138 | 149
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-USA: number analyzed (Participants) | 78 | 55 | 76 | 49 | 40 | 28 | 72 | 75 | 73 | 50 | 64
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 4-USA | 69 | 50 | 65 | 43 | 37 | 26 | 61 | 65 | 62 | 47 | 54
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru: number analyzed (Participants) | 1 | 40 | 0 | 5 | 40 | 54 | 8 | 15 | 15 | 20 | 22
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru | 1 | 38 | 0 | 5 | 38 | 51 | 8 | 15 | 15 | 17 | 22
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total: number analyzed (Participants) | 16 | 84 | 16 | 63 | 110 | 138 | 27 | 38 | 43 | 63 | 64
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total | 12 | 74 | 12 | 56 | 97 | 123 | 23 | 35 | 40 | 51 | 59
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA: number analyzed (Participants) | 15 | 44 | 16 | 58 | 70 | 84 | 19 | 23 | 28 | 43 | 42
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA | 11 | 36 | 12 | 51 | 59 | 72 | 15 | 20 | 25 | 34 | 37
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru: number analyzed (Participants) | 5 | 42 | 0 | 8 | 43 | 51 | 7 | 15 | 10 | 21 | 17
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru | 5 | 39 | 0 | 8 | 40 | 47 | 6 | 15 | 10 | 18 | 17
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total: number analyzed (Participants) | 18 | 92 | 12 | 74 | 125 | 139 | 29 | 35 | 26 | 71 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total | 13 | 80 | 9 | 64 | 109 | 123 | 26 | 34 | 24 | 59 | 46
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA: number analyzed (Participants) | 13 | 50 | 12 | 66 | 82 | 88 | 22 | 20 | 16 | 50 | 33
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA | 8 | 41 | 9 | 56 | 69 | 76 | 20 | 19 | 14 | 41 | 29
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 31 | 0 | 7 | 32 | 40 | 6 | 12 | 6 | 19 | 11
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-Peru | 5 | 27 | 0 | 6 | 28 | 35 | 5 | 12 | 6 | 15 | 11
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 98 | 20 | 23 | 19 | 55 | 33
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-Total | 11 | 52 | 10 | 38 | 66 | 84 | 19 | 22 | 19 | 43 | 32
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 58 | 14 | 11 | 13 | 36 | 22
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 4-USA | 6 | 25 | 10 | 32 | 38 | 49 | 14 | 10 | 13 | 28 | 21
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru: number analyzed (Participants) | 163 | 120 | 169 | 161 | 120 | 109 | 161 | 154 | 154 | 144 | 146
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru | 154 | 114 | 160 | 153 | 114 | 105 | 152 | 145 | 145 | 140 | 137
  SARS-CoV-2 S1 C His-50-N at Month 0-Total: number analyzed (Participants) | 335 | 242 | 337 | 262 | 201 | 182 | 320 | 315 | 315 | 273 | 284
  SARS-CoV-2 S1 C His-50-N at Month 0-Total | 300 | 216 | 302 | 236 | 181 | 167 | 283 | 279 | 278 | 252 | 251
  SARS-CoV-2 S1 C His-50-N at Month 0-USA: number analyzed (Participants) | 172 | 122 | 168 | 101 | 81 | 73 | 159 | 161 | 161 | 129 | 138
  SARS-CoV-2 S1 C His-50-N at Month 0-USA | 146 | 102 | 142 | 83 | 67 | 62 | 131 | 134 | 133 | 112 | 114
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru: number analyzed (Participants) | 134 | 97 | 140 | 132 | 96 | 88 | 133 | 125 | 130 | 119 | 122
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru | 125 | 91 | 131 | 123 | 90 | 83 | 125 | 116 | 121 | 113 | 113
  SARS-CoV-2 S1 C His-50-N at Month 2-Total: number analyzed (Participants) | 258 | 184 | 264 | 202 | 150 | 136 | 248 | 242 | 250 | 206 | 225
  SARS-CoV-2 S1 C His-50-N at Month 2-Total | 235 | 168 | 239 | 184 | 138 | 126 | 223 | 215 | 225 | 190 | 203
  SARS-CoV-2 S1 C His-50-N at Month 2-USA: number analyzed (Participants) | 124 | 87 | 124 | 70 | 54 | 48 | 115 | 117 | 120 | 87 | 103
  SARS-CoV-2 S1 C His-50-N at Month 2-USA | 110 | 77 | 108 | 61 | 48 | 43 | 98 | 99 | 104 | 77 | 90
  SARS-CoV-2 S1 C His-50-N at Month 4-Peru: number analyzed (Participants) | 109 | 83 | 114 | 107 | 82 | 75 | 109 | 102 | 108 | 95 | 104
  SARS-CoV-2 S1 C His-50-N at Month 4-Peru | 100 | 78 | 105 | 99 | 77 | 71 | 101 | 93 | 99 | 90 | 95
  SARS-CoV-2 S1 C His-50-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 103 | 181 | 177 | 181 | 145 | 168
  SARS-CoV-2 S1 C His-50-N at Month 4-Total | 168 | 127 | 169 | 141 | 113 | 97 | 160 | 156 | 161 | 136 | 149
  SARS-CoV-2 S1 C His-50-N at Month 4-USA: number analyzed (Participants) | 78 | 55 | 76 | 49 | 40 | 28 | 72 | 75 | 73 | 50 | 64
  SARS-CoV-2 S1 C His-50-N at Month 4-USA | 68 | 49 | 64 | 42 | 36 | 26 | 59 | 63 | 62 | 46 | 54
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru: number analyzed (Participants) | 6 | 49 | 0 | 8 | 49 | 60 | 8 | 15 | 15 | 25 | 23
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru | 6 | 46 | 0 | 7 | 46 | 55 | 8 | 15 | 15 | 20 | 23
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 96 | 157 | 176 | 38 | 43 | 43 | 85 | 74
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total | 17 | 101 | 15 | 81 | 136 | 150 | 34 | 38 | 39 | 65 | 66
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 88 | 108 | 116 | 30 | 28 | 28 | 60 | 51
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA | 11 | 55 | 15 | 74 | 90 | 95 | 26 | 23 | 24 | 45 | 43
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru: number analyzed (Participants) | 6 | 43 | 0 | 8 | 44 | 52 | 7 | 15 | 10 | 21 | 18
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru | 6 | 40 | 0 | 8 | 41 | 48 | 6 | 15 | 10 | 18 | 18
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 13 | 75 | 127 | 141 | 29 | 35 | 27 | 71 | 52
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total | 14 | 81 | 10 | 65 | 111 | 123 | 26 | 34 | 24 | 59 | 46
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA: number analyzed (Participants) | 13 | 50 | 13 | 67 | 83 | 89 | 22 | 20 | 17 | 50 | 34
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA | 8 | 41 | 10 | 57 | 70 | 75 | 20 | 19 | 14 | 41 | 28
  SARS-CoV-2 S1 C His-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 31 | 0 | 7 | 32 | 39 | 5 | 12 | 6 | 19 | 10
  SARS-CoV-2 S1 C His-50-Y at Month 4-Peru | 5 | 27 | 0 | 6 | 28 | 34 | 4 | 12 | 6 | 15 | 10
  SARS-CoV-2 S1 C His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 97 | 19 | 23 | 19 | 55 | 32
  SARS-CoV-2 S1 C His-50-Y at Month 4-Total | 10 | 51 | 9 | 37 | 65 | 81 | 18 | 22 | 17 | 42 | 29
  SARS-CoV-2 S1 C His-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 58 | 14 | 11 | 13 | 36 | 22
  SARS-CoV-2 S1 C His-50-Y at Month 4-USA | 5 | 24 | 9 | 31 | 37 | 47 | 14 | 10 | 11 | 27 | 19
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru: number analyzed (Participants) | 166 | 122 | 173 | 164 | 121 | 113 | 165 | 158 | 158 | 148 | 150
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru | 156 | 116 | 163 | 155 | 115 | 108 | 156 | 148 | 148 | 142 | 140
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 341 | 245 | 345 | 267 | 203 | 187 | 327 | 322 | 322 | 278 | 291
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total | 313 | 223 | 316 | 246 | 188 | 174 | 297 | 291 | 292 | 259 | 263
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA: number analyzed (Participants) | 175 | 123 | 172 | 103 | 82 | 74 | 162 | 164 | 164 | 130 | 141
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA | 157 | 107 | 153 | 91 | 73 | 66 | 141 | 143 | 144 | 117 | 123
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru: number analyzed (Participants) | 129 | 93 | 135 | 127 | 92 | 85 | 128 | 120 | 125 | 114 | 119
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru | 122 | 89 | 128 | 120 | 88 | 81 | 122 | 113 | 118 | 109 | 112
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 249 | 177 | 255 | 197 | 146 | 130 | 238 | 230 | 242 | 194 | 219
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total | 233 | 166 | 237 | 184 | 139 | 123 | 221 | 212 | 223 | 184 | 202
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA: number analyzed (Participants) | 120 | 84 | 120 | 70 | 54 | 45 | 110 | 110 | 117 | 80 | 100
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA | 111 | 77 | 109 | 64 | 51 | 42 | 99 | 99 | 105 | 75 | 90
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-Peru: number analyzed (Participants) | 102 | 77 | 106 | 99 | 76 | 70 | 102 | 94 | 100 | 89 | 97
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-Peru | 96 | 74 | 100 | 93 | 73 | 67 | 97 | 88 | 94 | 85 | 91
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-Total: number analyzed (Participants) | 176 | 129 | 178 | 146 | 114 | 95 | 170 | 165 | 170 | 136 | 158
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-Total | 163 | 122 | 163 | 135 | 109 | 90 | 155 | 150 | 155 | 129 | 144
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-USA: number analyzed (Participants) | 74 | 52 | 72 | 47 | 38 | 25 | 68 | 71 | 70 | 47 | 61
  SARS-CoV-2 S1S2 ECD His-50-N at Month 4-USA | 67 | 48 | 63 | 42 | 36 | 23 | 58 | 62 | 61 | 44 | 53
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 60 | 8 | 15 | 15 | 25 | 23
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru | 7 | 47 | 0 | 8 | 48 | 55 | 7 | 15 | 15 | 21 | 23
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 20 | 98 | 162 | 178 | 38 | 43 | 43 | 87 | 74
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total | 18 | 108 | 15 | 85 | 143 | 157 | 34 | 40 | 39 | 72 | 68
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA: number analyzed (Participants) | 17 | 69 | 20 | 89 | 110 | 118 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA | 11 | 61 | 15 | 77 | 95 | 102 | 27 | 25 | 24 | 51 | 45
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru: number analyzed (Participants) | 6 | 42 | 0 | 8 | 43 | 50 | 7 | 15 | 10 | 21 | 16
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru | 6 | 39 | 0 | 8 | 40 | 47 | 6 | 15 | 10 | 19 | 16
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 16 | 88 | 10 | 68 | 119 | 135 | 27 | 35 | 23 | 71 | 46
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total | 13 | 80 | 9 | 62 | 107 | 123 | 25 | 34 | 23 | 62 | 44
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA: number analyzed (Participants) | 10 | 46 | 10 | 60 | 76 | 85 | 20 | 20 | 13 | 50 | 30
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA | 7 | 41 | 9 | 54 | 67 | 76 | 19 | 19 | 13 | 43 | 28
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-Peru: number analyzed (Participants) | 4 | 29 | 0 | 7 | 30 | 36 | 4 | 12 | 6 | 17 | 9
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-Peru | 4 | 26 | 0 | 7 | 27 | 33 | 3 | 12 | 6 | 15 | 9
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-Total: number analyzed (Participants) | 12 | 59 | 10 | 42 | 74 | 93 | 18 | 23 | 18 | 52 | 30
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-Total | 9 | 50 | 9 | 37 | 63 | 82 | 17 | 22 | 17 | 43 | 28
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 30 | 10 | 35 | 44 | 57 | 14 | 11 | 12 | 35 | 21
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 4-USA | 5 | 24 | 9 | 30 | 36 | 49 | 14 | 10 | 11 | 28 | 19
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru: number analyzed (Participants) | 169 | 125 | 176 | 167 | 124 | 113 | 167 | 159 | 161 | 151 | 153
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru | 159 | 119 | 166 | 158 | 118 | 109 | 158 | 149 | 151 | 146 | 143
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total: number analyzed (Participants) | 345 | 249 | 349 | 271 | 207 | 187 | 330 | 324 | 326 | 282 | 295
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total | 313 | 227 | 317 | 249 | 192 | 175 | 298 | 291 | 292 | 264 | 264
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA: number analyzed (Participants) | 176 | 124 | 173 | 104 | 83 | 74 | 163 | 165 | 165 | 131 | 142
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA | 154 | 108 | 151 | 91 | 74 | 66 | 140 | 142 | 141 | 118 | 121
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru: number analyzed (Participants) | 134 | 97 | 139 | 131 | 96 | 88 | 132 | 124 | 129 | 118 | 122
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru | 125 | 92 | 130 | 123 | 91 | 84 | 124 | 115 | 120 | 113 | 113
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total: number analyzed (Participants) | 258 | 184 | 264 | 202 | 151 | 137 | 248 | 242 | 251 | 205 | 227
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total | 238 | 171 | 242 | 187 | 142 | 129 | 227 | 219 | 228 | 193 | 206
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA: number analyzed (Participants) | 124 | 87 | 125 | 71 | 55 | 49 | 116 | 118 | 122 | 87 | 105
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA | 113 | 79 | 112 | 64 | 51 | 45 | 103 | 104 | 108 | 80 | 93
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-Peru: number analyzed (Participants) | 110 | 83 | 115 | 108 | 82 | 75 | 109 | 103 | 109 | 96 | 104
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-Peru | 102 | 79 | 107 | 101 | 78 | 72 | 102 | 95 | 101 | 92 | 96
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-Total: number analyzed (Participants) | 189 | 139 | 192 | 158 | 123 | 103 | 182 | 178 | 183 | 146 | 169
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-Total | 172 | 130 | 173 | 145 | 116 | 98 | 164 | 160 | 164 | 139 | 151
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-USA: number analyzed (Participants) | 79 | 56 | 77 | 50 | 41 | 28 | 73 | 75 | 74 | 50 | 65
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 4-USA | 70 | 51 | 66 | 44 | 38 | 26 | 62 | 65 | 63 | 47 | 55
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 63 | 9 | 17 | 15 | 25 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru | 7 | 47 | 0 | 8 | 48 | 57 | 8 | 17 | 15 | 20 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 20 | 98 | 162 | 182 | 39 | 45 | 43 | 87 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total | 19 | 105 | 15 | 83 | 140 | 157 | 34 | 41 | 40 | 68 | 68
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA: number analyzed (Participants) | 17 | 69 | 20 | 89 | 110 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA | 12 | 58 | 15 | 75 | 92 | 100 | 26 | 24 | 25 | 48 | 45
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru: number analyzed (Participants) | 5 | 42 | 0 | 8 | 43 | 51 | 7 | 15 | 10 | 21 | 17
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru | 5 | 38 | 0 | 7 | 39 | 46 | 6 | 15 | 10 | 17 | 17
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 13 | 75 | 126 | 140 | 29 | 35 | 26 | 72 | 50
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total | 15 | 82 | 11 | 66 | 111 | 124 | 26 | 34 | 25 | 60 | 47
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA: number analyzed (Participants) | 14 | 51 | 13 | 67 | 83 | 89 | 22 | 20 | 16 | 51 | 33
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA | 10 | 44 | 11 | 59 | 72 | 78 | 20 | 19 | 15 | 43 | 30
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 32 | 0 | 7 | 33 | 40 | 6 | 12 | 6 | 19 | 11
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-Peru | 5 | 28 | 0 | 6 | 29 | 35 | 5 | 12 | 6 | 15 | 11
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 99 | 20 | 24 | 19 | 56 | 33
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-Total | 11 | 53 | 10 | 38 | 67 | 85 | 19 | 23 | 19 | 44 | 32
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 59 | 14 | 12 | 13 | 37 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 4-USA | 6 | 25 | 10 | 32 | 38 | 50 | 14 | 11 | 13 | 29 | 21
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru: number analyzed (Participants) | 140 | 101 | 142 | 137 | 101 | 87 | 134 | 128 | 127 | 121 | 119
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru | 136 | 99 | 138 | 133 | 99 | 86 | 130 | 124 | 123 | 120 | 115
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total: number analyzed (Participants) | 251 | 182 | 252 | 205 | 156 | 128 | 240 | 231 | 225 | 204 | 203
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total | 236 | 173 | 236 | 193 | 150 | 125 | 224 | 213 | 210 | 197 | 190
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA: number analyzed (Participants) | 111 | 81 | 110 | 68 | 55 | 41 | 106 | 103 | 98 | 83 | 84
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA | 100 | 74 | 98 | 60 | 51 | 39 | 94 | 89 | 87 | 77 | 75
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru: number analyzed (Participants) | 132 | 95 | 138 | 130 | 94 | 87 | 131 | 123 | 128 | 117 | 121
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru | 123 | 89 | 129 | 121 | 88 | 82 | 123 | 114 | 119 | 111 | 112
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total: number analyzed (Participants) | 250 | 177 | 257 | 198 | 146 | 132 | 241 | 234 | 242 | 201 | 220
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total | 228 | 161 | 232 | 180 | 134 | 122 | 217 | 207 | 218 | 186 | 198
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA: number analyzed (Participants) | 118 | 82 | 119 | 68 | 52 | 45 | 110 | 111 | 114 | 84 | 99
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA | 105 | 72 | 103 | 59 | 46 | 40 | 94 | 93 | 99 | 75 | 86
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-Peru: number analyzed (Participants) | 110 | 83 | 115 | 108 | 82 | 75 | 109 | 103 | 109 | 96 | 104
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-Peru | 103 | 79 | 108 | 101 | 78 | 72 | 103 | 96 | 102 | 92 | 97
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-Total: number analyzed (Participants) | 188 | 138 | 191 | 157 | 122 | 103 | 181 | 178 | 182 | 146 | 168
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-Total | 171 | 128 | 171 | 143 | 114 | 98 | 162 | 158 | 164 | 138 | 151
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-USA: number analyzed (Participants) | 78 | 55 | 76 | 49 | 40 | 28 | 72 | 75 | 73 | 50 | 64
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 4-USA | 68 | 49 | 63 | 42 | 36 | 26 | 59 | 62 | 62 | 46 | 54
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru: number analyzed (Participants) | 2 | 41 | 0 | 5 | 41 | 55 | 8 | 14 | 15 | 21 | 23
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru | 2 | 39 | 0 | 5 | 39 | 52 | 8 | 14 | 15 | 18 | 23
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total: number analyzed (Participants) | 17 | 86 | 16 | 63 | 112 | 140 | 28 | 37 | 43 | 64 | 65
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total | 11 | 74 | 11 | 54 | 97 | 122 | 23 | 34 | 37 | 50 | 57
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA: number analyzed (Participants) | 15 | 45 | 16 | 58 | 71 | 85 | 20 | 23 | 28 | 43 | 42
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA | 9 | 35 | 11 | 49 | 58 | 70 | 15 | 20 | 22 | 32 | 34
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru: number analyzed (Participants) | 6 | 43 | 0 | 8 | 44 | 51 | 7 | 15 | 10 | 21 | 17
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru | 6 | 40 | 0 | 8 | 41 | 47 | 6 | 15 | 10 | 18 | 17
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 92 | 12 | 71 | 123 | 137 | 28 | 35 | 27 | 68 | 49
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total | 13 | 80 | 9 | 61 | 107 | 119 | 24 | 34 | 23 | 55 | 43
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA: number analyzed (Participants) | 13 | 49 | 12 | 63 | 79 | 86 | 21 | 20 | 17 | 47 | 32
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA | 7 | 40 | 9 | 53 | 66 | 72 | 18 | 19 | 13 | 37 | 26
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-Peru: number analyzed (Participants) | 5 | 32 | 0 | 7 | 33 | 40 | 6 | 12 | 6 | 19 | 11
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-Peru | 5 | 29 | 0 | 7 | 30 | 36 | 5 | 12 | 6 | 16 | 11
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 98 | 20 | 23 | 19 | 55 | 33
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-Total | 9 | 52 | 9 | 37 | 66 | 82 | 18 | 22 | 16 | 42 | 29
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-USA: number analyzed (Participants) | 8 | 31 | 10 | 37 | 46 | 58 | 14 | 11 | 13 | 36 | 22
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 4-USA | 4 | 23 | 9 | 30 | 36 | 46 | 13 | 10 | 10 | 26 | 18

47. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG1) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG1) at Visit 1, 2, 3, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2, 4
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
MFI
  2019-nCoV S/293F-1000-N at Month 0-Total: number analyzed (Participants) | 264 | 190 | 268 | 218 | 162 | 139 | 256 | 245 | 241 | 217 | 219
  2019-nCoV S/293F-1000-N at Month 0-Total | 21989.8 [7432.8 to 22000] | 21924.8 [5983.1 to 22000] | 21849.4 [7671.6 to 22000] | 22000 [8074.5 to 22000] | 22000 [8187.4 to 22000] | 22000 [8304.9 to 22000] | 21664.4 [7036.2 to 22000] | 20217 [5081 to 22000] | 21972.8 [6757 to 22000] | 20312 [6287 to 22000] | 22000 [7581.1 to 22000]
  2019-nCoV S/293F-1000-N at Month 2-Total: number analyzed (Participants) | 253 | 179 | 261 | 200 | 148 | 131 | 243 | 237 | 245 | 201 | 220
  2019-nCoV S/293F-1000-N at Month 2-Total | 9624.5 [2984.2 to 20483.8] | 9478 [3120.6 to 20452.5] | 9065.8 [2876.8 to 20056.2] | 10137.4 [2844.3 to 22000] | 10664.6 [2844.3 to 22000] | 7601 [2509.1 to 20175] | 8898.8 [2675.8 to 20282.1] | 7601 [2010 to 19418] | 9065.8 [2711.8 to 20421.2] | 7577 [2621.2 to 18828.5] | 8894.8 [2522.9 to 20959.9]
  2019-nCoV S/293F-1000-N at Month 4-Total: number analyzed (Participants) | 189 | 139 | 192 | 158 | 123 | 103 | 182 | 178 | 183 | 146 | 169
  2019-nCoV S/293F-1000-N at Month 4-Total | 4279 [1288 to 14394.3] | 4413 [1514.2 to 14348] | 3677.9 [1125.2 to 14200.1] | 4408.1 [1408 to 14901.8] | 4763.8 [1662.5 to 15050.4] | 3660 [1159.1 to 14274] | 4158 [1054.6 to 14581.6] | 3196.9 [989.9 to 12670.5] | 3695.8 [1159.1 to 14837] | 3414.9 [1146.9 to 13275.6] | 3660 [1096.8 to 14966.5]
  2019-nCoV S/293F-1000-Y at Month 0-Total: number analyzed (Participants) | 20 | 94 | 16 | 66 | 122 | 145 | 28 | 39 | 43 | 67 | 65
  2019-nCoV S/293F-1000-Y at Month 0-Total | 4569.9 [558.9 to 13484.9] | 16577.6 [5504.6 to 22000] | 1313.2 [195.2 to 7612.6] | 10749.1 [2478.1 to 22000] | 14683.4 [4002.6 to 22000] | 16814.5 [4307.8 to 22000] | 9277.6 [1466.2 to 22000] | 22000 [10521.1 to 22000] | 13720.2 [3015 to 22000] | 22000 [4025.2 to 22000] | 13720.2 [4110.8 to 22000]
  2019-nCoV S/293F-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 11 | 72 | 124 | 141 | 29 | 35 | 27 | 71 | 52
  2019-nCoV S/293F-1000-Y at Month 2-Total | 2711.8 [129.6 to 6004.5] | 6956.8 [1850 to 16844.2] | 759 [182.9 to 5334.6] | 5077.1 [1741.8 to 13177.6] | 6829.5 [1988.8 to 15928.2] | 9271.5 [2747 to 19418] | 8553.8 [1792.2 to 15764.8] | 12426.2 [6736.9 to 21241.9] | 4956.2 [1901.1 to 16606.4] | 11437.8 [2336.2 to 20313.4] | 7388.8 [2720.2 to 17521.3]
  2019-nCoV S/293F-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 99 | 20 | 24 | 19 | 56 | 33
  2019-nCoV S/293F-1000-Y at Month 4-Total | 958.5 [261.5 to 1857.2] | 2272.5 [554.8 to 13357.6] | 2031.9 [764 to 5144.6] | 1777 [524.5 to 8249.4] | 2265 [608.2 to 11582.6] | 3382.2 [999.5 to 13315.5] | 2125.2 [1665.2 to 5108.5] | 8224.2 [2391.2 to 21245.9] | 2586.8 [956.9 to 5435.5] | 4913.5 [930.2 to 15008.4] | 3382.2 [1415 to 9555.5]
  229E-RBD-50-N at Month 0-Total: number analyzed (Participants) | 245 | 179 | 244 | 200 | 153 | 125 | 234 | 221 | 220 | 201 | 199
  229E-RBD-50-N at Month 0-Total | 5540 [3473 to 8258.8] | 5035.8 [3318.1 to 8428.1] | 5623.4 [3593.2 to 8113.5] | 5836.9 [3609.8 to 8493.4] | 5609 [3440.2 to 8486.8] | 5818.2 [3744 to 8513.5] | 5574.5 [3448.4 to 8262.9] | 5444.8 [3314.8 to 8098.2] | 5766.9 [3392.8 to 8260.1] | 5536.8 [3678.8 to 8098.2] | 5775.5 [3456.6 to 8520]
  229E-RBD-50-N at Month 2-Total: number analyzed (Participants) | 242 | 173 | 247 | 189 | 139 | 131 | 234 | 232 | 236 | 194 | 212
  229E-RBD-50-N at Month 2-Total | 5174.8 [2927.1 to 8040.9] | 4738.2 [2894.5 to 7856] | 5268.5 [3002 to 8012.8] | 5494 [3159.8 to 8219.2] | 4801.8 [2921.6 to 8006] | 5268.5 [3370.4 to 7887.1] | 5279 [2945 to 8037.5] | 4890.2 [2902.9 to 7926.7] | 5057.6 [2969.5 to 7946.4] | 4936.8 [2991.9 to 7896.9] | 5174.8 [3272.6 to 7974.5]
  229E-RBD-50-N at Month 4-Total: number analyzed (Participants) | 168 | 126 | 171 | 139 | 110 | 91 | 164 | 160 | 163 | 130 | 152
  229E-RBD-50-N at Month 4-Total | 6282.2 [3977.9 to 8734.1] | 6242.8 [3980.8 to 8614.3] | 6289 [3985.2 to 9007.6] | 6379.5 [4149.4 to 9789] | 6274 [4094.1 to 9642.9] | 6289 [4307.6 to 8392.5] | 6334.2 [4053.5 to 8639.6] | 6275 [3951.9 to 8639.6] | 6289 [4030.2 to 8793.2] | 6439.2 [4094.1 to 8614.3] | 6282.2 [4053.1 to 8734.1]
  229E-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 15 | 81 | 16 | 60 | 107 | 135 | 26 | 39 | 40 | 59 | 61
  229E-RBD-50-Y at Month 0-Total | 5227.2 [2054.2 to 5914.5] | 5877 [3827.8 to 7704.2] | 3361.8 [1933.2 to 6372.1] | 4230.4 [2810.8 to 6882.3] | 5522.2 [3367.8 to 7766.8] | 5418.8 [3251.2 to 7770.5] | 5256 [3314.4 to 6943.9] | 5786.5 [3598.8 to 7804.5] | 5288 [3688.6 to 7387.4] | 5449.5 [2743.6 to 8031.1] | 5284.8 [3283 to 7182.5]
  229E-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 88 | 14 | 72 | 122 | 130 | 27 | 29 | 25 | 67 | 49
  229E-RBD-50-Y at Month 2-Total | 4083.2 [3500 to 5991.9] | 5584.2 [3557.1 to 7987.2] | 3677.4 [2271 to 4456] | 4425.9 [2664.4 to 6593.4] | 5078.5 [3219.3 to 7872.6] | 4986.8 [2838.2 to 7947.7] | 4654.2 [2924.1 to 6766] | 5982 [4185.8 to 7856] | 4939.2 [2564.2 to 7112.2] | 5106.8 [2686.2 to 8144.1] | 4693.2 [2564.2 to 7217]
  229E-RBD-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 55 | 10 | 42 | 71 | 90 | 17 | 21 | 18 | 51 | 29
  229E-RBD-50-Y at Month 4-Total | 6172.5 [4225.2 to 7904.2] | 6873 [4187.8 to 9007.6] | 5991.4 [3176.1 to 6940.4] | 5991.4 [3157.6 to 7880.9] | 6451.2 [3748.5 to 8392.5] | 6235.8 [3804.7 to 9948.3] | 4989 [3787.8 to 9733.8] | 6878 [5495.2 to 10318.8] | 5978.9 [3714.5 to 8065.7] | 6014.2 [3782.4 to 9913.6] | 6198 [3624 to 8119.5]
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 318 | 229 | 321 | 246 | 188 | 171 | 307 | 299 | 300 | 259 | 276
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total | 14162.9 [7994.5 to 21650.9] | 14355 [8411.5 to 21795] | 13899 [7734.8 to 21510.5] | 14104.4 [8279 to 21412] | 14305.4 [8220.8 to 21459.3] | 16171.8 [9845.8 to 22000] | 14013.5 [8116.6 to 21986.4] | 14355 [8407.5 to 21893.4] | 14162.9 [8040 to 21979.6] | 14355 [8204 to 22000] | 14321.1 [8362 to 22000]
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 245 | 176 | 250 | 192 | 142 | 132 | 236 | 234 | 238 | 196 | 213
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total | 9586.8 [5500.8 to 15912.5] | 9248.6 [5464.1 to 14802.1] | 9590.6 [5548.9 to 15837] | 9633 [5769.9 to 15966] | 9108.8 [5308.2 to 14737.4] | 11154.8 [6583.8 to 16753] | 9652.1 [5709.2 to 16035.9] | 9613.6 [5558.7 to 15992.8] | 9574.4 [5548.9 to 15992.8] | 9677.5 [5735.5 to 16035.9] | 9798 [6045 to 16144]
  HCoV-229E S1S2 ECD His-50-N at Month 4-Total: number analyzed (Participants) | 181 | 135 | 184 | 151 | 119 | 99 | 174 | 172 | 176 | 141 | 162
  HCoV-229E S1S2 ECD His-50-N at Month 4-Total | 10361.8 [6110.5 to 15266.8] | 9486 [6122.4 to 14005.1] | 10086.5 [6078.1 to 15237.9] | 10455.5 [6122.4 to 15026.1] | 9645.5 [6122.4 to 14005.1] | 10725.5 [7237.2 to 17708.5] | 10408.6 [6251.1 to 16007.9] | 10458.6 [6351.4 to 15892.9] | 9838 [6078.1 to 15237.9] | 10148.5 [6257.5 to 15266.8] | 10458.6 [6251.1 to 16007.9]
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 113 | 21 | 96 | 154 | 171 | 35 | 43 | 42 | 83 | 66
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total | 10434.5 [6422.4 to 15676.5] | 12464.8 [6964 to 21070.2] | 13250.5 [9134.8 to 22000] | 13181 [6074.3 to 22000] | 13155.8 [7391.9 to 21785.3] | 11441.5 [6040.8 to 19863.4] | 12464.8 [6699.1 to 19873.2] | 10571.5 [3394.6 to 17391.2] | 11550.1 [6209.4 to 17355.2] | 11759.5 [6604.9 to 19733.8] | 11550.1 [5329.9 to 18223.3]
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 18 | 87 | 13 | 71 | 121 | 131 | 27 | 29 | 25 | 67 | 50
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total | 9540.6 [7691.7 to 12558.4] | 9870.5 [6493.5 to 16509.5] | 8755.8 [7061.2 to 16964.2] | 9129.8 [5404 to 14616.2] | 9817.5 [6491.8 to 16085] | 8861.8 [5176.6 to 14424] | 8364.2 [4660.8 to 13029.8] | 9246 [5611 to 14104.8] | 9662.2 [5779.2 to 13466.2] | 9195.8 [5418.9 to 14914.5] | 8986 [4097.8 to 12570.7]
  HCoV-229E S1S2 ECD His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 59 | 10 | 43 | 75 | 95 | 20 | 22 | 18 | 53 | 32
  HCoV-229E S1S2 ECD His-50-Y at Month 4-Total | 9386.8 [7725.8 to 13002.2] | 12195 [6172.5 to 17234.1] | 12681.8 [7818.5 to 14691.6] | 9651.5 [6075 to 16727] | 10725.5 [6172.5 to 17234.1] | 8857.8 [5071.8 to 13845.6] | 9061.5 [3213.4 to 12950.6] | 7908 [5275.7 to 12630.5] | 12775.5 [7253.1 to 15017.1] | 10489 [5023.8 to 14830.8] | 8486.1 [5120.7 to 13096.9]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 317 | 229 | 320 | 246 | 188 | 171 | 306 | 298 | 300 | 259 | 276
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total | 15344 [8541.5 to 22000] | 15952.5 [8730.8 to 22000] | 15079 [8305.9 to 22000] | 15229.8 [8748.2 to 22000] | 15612.2 [9132.9 to 22000] | 15373.5 [8777.1 to 22000] | 14854.8 [8136.1 to 22000] | 15364.2 [8301.6 to 22000] | 15128.1 [8269.6 to 22000] | 15053.5 [8476.2 to 22000] | 15128.1 [8648.3 to 22000]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 244 | 175 | 250 | 192 | 142 | 131 | 236 | 233 | 238 | 196 | 213
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total | 13900.9 [8117.6 to 20949.1] | 14306 [7868.5 to 20955.6] | 13531.1 [7893 to 21146.7] | 13900.9 [7869.1 to 21318.1] | 13900.9 [7174.1 to 20962.2] | 13272.5 [8844.9 to 19898.2] | 13385.6 [7946 to 20937.8] | 13674.5 [8254.5 to 21485.2] | 13636.8 [7912.5 to 21278] | 13289.4 [8231.2 to 18974.3] | 13599 [7962.8 to 20936.2]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 103 | 180 | 178 | 181 | 145 | 167
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 4-Total | 13428.8 [7426.6 to 21301.6] | 13633.4 [7487.9 to 21319.9] | 12463.2 [7149.4 to 20989.4] | 12836.9 [7083.6 to 21079.9] | 12836.9 [7487.9 to 21203.3] | 13838 [7546.5 to 22000] | 12836.9 [7391.4 to 20993.3] | 13915 [8153.1 to 21358.9] | 12878 [7098.2 to 21338.2] | 12795.8 [7302.8 to 21018.2] | 12878 [7200.5 to 20934.1]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 112 | 21 | 95 | 153 | 170 | 35 | 43 | 41 | 82 | 65
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total | 10845.4 [3583.1 to 19334.5] | 13251.2 [6947.3 to 21628.1] | 10994 [4651 to 22000] | 14726.2 [7111.8 to 22000] | 14590.5 [7245.2 to 22000] | 14590.8 [7128.4 to 21713.1] | 16454 [8119.5 to 22000] | 12192.5 [6866.1 to 19986.5] | 13531.5 [7623 to 19807.2] | 14860.1 [6737.5 to 21933.6] | 13531.5 [6395.5 to 21852]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 88 | 13 | 71 | 121 | 132 | 27 | 30 | 25 | 67 | 50
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total | 9758 [5391.1 to 19430.1] | 12312 [8227.7 to 20364.9] | 11412.8 [7895.8 to 18992.5] | 13072.5 [7929.2 to 19438] | 13072.5 [8254.5 to 20084.5] | 14208.1 [6780.3 to 21527.6] | 14306 [5419.5 to 21651] | 11415.8 [4406.6 to 17363.2] | 10813 [6863 to 17054] | 16129.8 [6936.6 to 22000] | 12770.5 [6104.6 to 21566.4]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 97 | 20 | 22 | 19 | 55 | 33
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 4-Total | 10934.5 [6837 to 14251.5] | 12053.1 [6855.2 to 19187.6] | 17832.9 [12435.7 to 20171.8] | 12901.2 [8906.9 to 19788.9] | 12901.2 [6855.2 to 20640.8] | 12048.5 [6837 to 20820.8] | 13150 [5131.4 to 19789.8] | 8077.2 [6668.9 to 15701.9] | 12795.8 [9247.1 to 18014.5] | 13440.5 [8778.4 to 20358.9] | 12795.8 [8737.2 to 20902.8]
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 318 | 229 | 321 | 246 | 188 | 171 | 307 | 300 | 299 | 259 | 275
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total | 1217.2 [36.1 to 2830.1] | 1260.8 [88.8 to 2830.2] | 1197.8 [50 to 2784.2] | 1104.8 [1 to 2667.9] | 1088.1 [1 to 2720.4] | 1323 [375.4 to 2953.1] | 1273.5 [87.5 to 2885.5] | 1356.9 [245.1 to 3060.4] | 1242.5 [56.4 to 2830] | 1319.2 [240 to 2885.5] | 1261.2 [94 to 2751.9]
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 226 | 166 | 227 | 175 | 132 | 123 | 216 | 213 | 216 | 181 | 195
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total | 1679.1 [473.9 to 3929.6] | 1679.1 [473.9 to 3960.1] | 1675.2 [475.2 to 3784.4] | 1527.8 [464.5 to 3498.5] | 1478.8 [408.4 to 3505.9] | 1820 [668.6 to 4187.6] | 1741.6 [474.3 to 4184.8] | 1897 [602 to 4211.8] | 1664.5 [475.4 to 3834.2] | 1830.2 [602 to 4081.8] | 1727.2 [578.4 to 3784.4]
  HCoV-NL63 S1S2 ECD His-50-N at Month 4-Total: number analyzed (Participants) | 181 | 135 | 184 | 151 | 119 | 99 | 174 | 172 | 176 | 141 | 162
  HCoV-NL63 S1S2 ECD His-50-N at Month 4-Total | 1363.5 [621.2 to 2960.8] | 1333 [685.6 to 2722.2] | 1394.2 [634.1 to 2856.8] | 1363.5 [654.6 to 2714.9] | 1411 [743.1 to 2659.5] | 1552.5 [812.4 to 2903.1] | 1545.6 [654.3 to 3009.9] | 1562.5 [733.6 to 3075.3] | 1335.9 [621.1 to 2748.6] | 1552.5 [730.8 to 2845.5] | 1335.9 [642.9 to 2813.2]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 113 | 21 | 96 | 154 | 171 | 35 | 42 | 43 | 83 | 67
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total | 2299.1 [1198.5 to 3590] | 1510 [158.8 to 2889.2] | 2677.2 [2077.2 to 6059.5] | 1957.6 [249.6 to 4215.7] | 1645.6 [247.2 to 3436.8] | 1120.5 [1 to 2830] | 1393.8 [280.5 to 2859.8] | 127.5 [1 to 2085.1] | 1949 [304.4 to 3190.2] | 1010.2 [1 to 2833.9] | 1741.8 [43.6 to 3475.1]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 13 | 73 | 12 | 64 | 107 | 116 | 23 | 26 | 23 | 58 | 44
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total | 3012.5 [1207.8 to 4247.8] | 2125.8 [756.5 to 3926.8] | 4362.1 [2866.1 to 5211.4] | 3182.1 [869.6 to 4806.2] | 2238.2 [761.4 to 4315.1] | 1452.4 [263.6 to 3797] | 1430 [837.9 to 3048.8] | 762.5 [1 to 2576] | 3515 [1013.8 to 4724.4] | 1267.1 [210.3 to 3486.1] | 1864.6 [15.4 to 4528.7]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 59 | 10 | 43 | 75 | 95 | 20 | 22 | 18 | 53 | 32
  HCoV-NL63 S1S2 ECD His-50-Y at Month 4-Total | 2059.2 [1473.2 to 3659.5] | 1934.2 [630 to 3356.1] | 3604.2 [1965.5 to 4232.3] | 2059.2 [621.6 to 3999.8] | 1572.5 [619.4 to 3487.2] | 1301 [593.9 to 3029.5] | 1171.2 [621.4 to 2791.1] | 717.8 [462.6 to 1925.3] | 2880.2 [2152.4 to 4232.3] | 1123 [583.8 to 3066.2] | 2445.6 [692.4 to 3525.1]
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 318 | 229 | 321 | 246 | 188 | 171 | 307 | 299 | 300 | 259 | 276
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total | 22000 [16980.8 to 22000] | 22000 [17027.2 to 22000] | 22000 [16922.8 to 22000] | 22000 [16906.6 to 22000] | 22000 [17092.6 to 22000] | 22000 [18309.2 to 22000] | 22000 [16892.4 to 22000] | 22000 [17177.6 to 22000] | 22000 [16620.8 to 22000] | 22000 [18468.4 to 22000] | 22000 [16947.5 to 22000]
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 245 | 177 | 250 | 193 | 143 | 132 | 238 | 234 | 238 | 198 | 214
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total | 22000 [16149 to 22000] | 22000 [16274.5 to 22000] | 22000 [15539.4 to 22000] | 22000 [15276 to 22000] | 22000 [15363.2 to 22000] | 22000 [17560.4 to 22000] | 22000 [15539.4 to 22000] | 22000 [15891.9 to 22000] | 22000 [15539.4 to 22000] | 22000 [16459.8 to 22000] | 22000 [16261.9 to 22000]
  HCoV-OC43 S1S2 ECD His-50-N at Month 4-Total: number analyzed (Participants) | 184 | 135 | 187 | 153 | 119 | 102 | 178 | 176 | 178 | 144 | 164
  HCoV-OC43 S1S2 ECD His-50-N at Month 4-Total | 22000 [13984.4 to 22000] | 21328.8 [14838.8 to 22000] | 21915.8 [13366.9 to 22000] | 21542 [13396.5 to 22000] | 21215.8 [14371.8 to 22000] | 22000 [13789.6 to 22000] | 22000 [13752.4 to 22000] | 22000 [13775.9 to 22000] | 21464.1 [13352.1 to 22000] | 22000 [13715.4 to 22000] | 21464.1 [13381.7 to 22000]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 113 | 21 | 96 | 154 | 171 | 35 | 43 | 42 | 83 | 66
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total | 21827.4 [11741.1 to 22000] | 21722.8 [16631.5 to 22000] | 22000 [16126.2 to 22000] | 22000 [16863.9 to 22000] | 22000 [16671 to 22000] | 22000 [14793.8 to 22000] | 22000 [19158.1 to 22000] | 21957 [14654.5 to 22000] | 22000 [19182.1 to 22000] | 21481.5 [12894.1 to 22000] | 22000 [16189.2 to 22000]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 87 | 14 | 71 | 121 | 132 | 26 | 30 | 26 | 66 | 50
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total | 21122.2 [6817.9 to 22000] | 22000 [13111.4 to 22000] | 22000 [14191.8 to 22000] | 22000 [16294.8 to 22000] | 22000 [15806.2 to 22000] | 22000 [12757.6 to 22000] | 22000 [12896.1 to 22000] | 22000 [9418.6 to 22000] | 22000 [14486.9 to 22000] | 22000 [12234.4 to 22000] | 22000 [12669.7 to 22000]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 95 | 19 | 21 | 19 | 53 | 33
  HCoV-OC43 S1S2 ECD His-50-Y at Month 4-Total | 21542 [9215.2 to 22000] | 22000 [11375.4 to 22000] | 22000 [19783.4 to 22000] | 22000 [14339.1 to 22000] | 22000 [12813.2 to 22000] | 21072.5 [13772.6 to 22000] | 20669.2 [14014.9 to 22000] | 19283 [13732.2 to 22000] | 22000 [14838.8 to 22000] | 21188.5 [14041.5 to 22000] | 22000 [14045.2 to 22000]
  HKU1-RBD-50-N at Month 0-Total: number analyzed (Participants) | 244 | 178 | 246 | 201 | 152 | 126 | 237 | 223 | 221 | 202 | 201
  HKU1-RBD-50-N at Month 0-Total | 4417.8 [2746.1 to 6576.1] | 4383.6 [2775.2 to 6561.8] | 4546.1 [2765.1 to 6857.2] | 4850.5 [2905.2 to 7278] | 4692.8 [2974.2 to 7264.4] | 5022.9 [3345.5 to 8375.9] | 4383.2 [2761.2 to 6568.8] | 4653.8 [2743.5 to 6942.6] | 4315 [2738.2 to 6761] | 4788.8 [2897.6 to 7145.5] | 4315 [2776.8 to 7037.5]
  HKU1-RBD-50-N at Month 2-Total: number analyzed (Participants) | 239 | 170 | 244 | 187 | 137 | 130 | 229 | 227 | 234 | 190 | 210
  HKU1-RBD-50-N at Month 2-Total | 4034.5 [1986.9 to 5865.8] | 4248.2 [2262.9 to 5911.7] | 4042.5 [2044.9 to 6017.1] | 4372 [2817.6 to 6127.2] | 4358.2 [2854.8 to 6138.5] | 4139.1 [2557.3 to 6591.2] | 4112.5 [2055.8 to 6024.2] | 4050.5 [2009 to 6019.5] | 4042.5 [1953.6 to 5883.4] | 4042.5 [2023.3 to 6037.8] | 4042.5 [2023.3 to 5823.9]
  HKU1-RBD-50-N at Month 4-Total: number analyzed (Participants) | 163 | 122 | 167 | 136 | 107 | 88 | 159 | 155 | 160 | 126 | 149
  HKU1-RBD-50-N at Month 4-Total | 5357.8 [2918 to 7899.5] | 5541.8 [3507.6 to 8396.4] | 5383.2 [3186.5 to 8259.6] | 5495.5 [3426.4 to 8225.7] | 5584.8 [3833.5 to 8528.8] | 5370.6 [3426.4 to 8367.6] | 5373 [3051.5 to 8064.2] | 5055.8 [2913.6 to 8272.2] | 5228.9 [2941.2 to 8127] | 5383.4 [3280.9 to 8084.4] | 5277.8 [3107.8 to 8194.5]
  HKU1-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 18 | 84 | 16 | 61 | 110 | 136 | 25 | 39 | 41 | 60 | 61
  HKU1-RBD-50-Y at Month 0-Total | 4014.5 [1340.1 to 5740.2] | 4322.4 [2267.9 to 6536.6] | 3121.6 [1741.8 to 4286.8] | 3371 [1201.2 to 4831.2] | 3816.2 [1881.8 to 5827.6] | 3808.2 [2207.6 to 5560.6] | 3781.8 [1995.2 to 5438] | 3517.2 [2284.6 to 5247.6] | 4487.5 [2625 to 5996.5] | 3514.5 [1768.2 to 5308.8] | 4487.5 [2497.2 to 6027.5]
  HKU1-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 17 | 86 | 12 | 69 | 119 | 126 | 27 | 29 | 22 | 66 | 46
  HKU1-RBD-50-Y at Month 2-Total | 3942.5 [1654.8 to 6107] | 3638.5 [1545.8 to 5786.7] | 2232.6 [1599.6 to 4732.1] | 2740.8 [1434 to 4985] | 3377.5 [1529 to 5631.6] | 3904.6 [1762.5 to 5503.4] | 3206.8 [1463.9 to 4969.1] | 3692.8 [1885.5 to 5108.5] | 3929.6 [2085.7 to 5930.9] | 3819.8 [1925.7 to 5725] | 3929.6 [1840.6 to 6738.3]
  HKU1-RBD-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 54 | 9 | 40 | 69 | 88 | 17 | 21 | 16 | 50 | 27
  HKU1-RBD-50-Y at Month 4-Total | 5655.8 [3042.5 to 8611.8] | 4234.1 [2646.6 to 6917.3] | 3042.5 [2783 to 5575.8] | 3923.8 [2481.8 to 7135.1] | 4078 [2576.5 to 7010.5] | 5343.1 [2780.5 to 7547.3] | 4047 [2234 to 8611.8] | 5655.8 [4656.2 to 6671] | 6419.4 [3050 to 7731.9] | 4933.5 [2775.5 to 8353.4] | 5759.2 [2756.6 to 7543.6]
  NL63-RBD-50-N at Month 0-Total: number analyzed (Participants) | 245 | 180 | 246 | 203 | 154 | 128 | 238 | 224 | 223 | 203 | 203
  NL63-RBD-50-N at Month 0-Total | 11600.8 [8579.2 to 16044.8] | 11438.5 [8578.4 to 16118.8] | 11798.5 [8604.9 to 16323.5] | 11690 [8630.5 to 15990.8] | 11552.5 [8604.9 to 15991.8] | 12737 [9631.6 to 16947.6] | 11934.4 [8766.1 to 16323.5] | 12039.9 [8746.9 to 16474.7] | 11325 [8483.4 to 15863.2] | 12258.5 [9282.1 to 16751.5] | 11577 [8577.6 to 16306.2]
  NL63-RBD-50-N at Month 2-Total: number analyzed (Participants) | 246 | 177 | 251 | 193 | 143 | 133 | 238 | 236 | 239 | 198 | 214
  NL63-RBD-50-N at Month 2-Total | 14274.4 [9800.2 to 17933.1] | 14453.2 [10202 to 17954.2] | 14451 [9913.2 to 18514.5] | 14451 [10485.8 to 18706] | 14572.8 [10482.1 to 18011.6] | 14715 [10478.5 to 18309.5] | 14500.8 [10190.8 to 18212.8] | 14500.8 [10359.3 to 18272.9] | 14233.2 [9725.5 to 18003.1] | 14537.2 [10434 to 18795.6] | 14315.5 [9904.7 to 17844]
  NL63-RBD-50-N at Month 4-Total: number analyzed (Participants) | 186 | 138 | 189 | 155 | 122 | 102 | 179 | 176 | 180 | 144 | 166
  NL63-RBD-50-N at Month 4-Total | 16414.2 [12580.9 to 19445.1] | 16306.5 [13066.1 to 19400] | 16447.5 [12503.2 to 19669] | 16602.5 [13493.2 to 19859] | 16491.6 [13475.5 to 19451.8] | 16491.6 [13385.2 to 19765.3] | 16381 [12521.4 to 19641.5] | 16491.6 [12923.2 to 19848.9] | 16171.4 [12404.4 to 19110] | 16547.5 [13296.8 to 20137.7] | 16171.4 [12436.3 to 19400]
  NL63-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 18 | 83 | 17 | 60 | 109 | 135 | 25 | 39 | 40 | 60 | 60
  NL63-RBD-50-Y at Month 0-Total | 13903.1 [12099.9 to 16639.2] | 12877.8 [9393.5 to 16104.2] | 13636.2 [9850 to 14738.5] | 12419.9 [8924.6 to 16561.6] | 12258.5 [8996 to 16271.8] | 11313 [8231.9 to 15137.6] | 10177 [7687 to 14040.5] | 11280.8 [8628.9 to 13364.6] | 13838.4 [11187.8 to 16813.8] | 9958.9 [7794.7 to 14416.5] | 12831.8 [9190.8 to 15914.4]
  NL63-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 88 | 14 | 72 | 122 | 132 | 27 | 29 | 26 | 67 | 51
  NL63-RBD-50-Y at Month 2-Total | 15792.8 [13948.6 to 20541.5] | 14215.4 [9762.2 to 19158.4] | 14352.6 [11602.3 to 15600.5] | 14352.6 [9472.9 to 17838.1] | 14201.5 [9538.2 to 18307.4] | 13960.9 [9762.2 to 18030.9] | 13571.2 [9980.9 to 17495.4] | 13393.8 [8592.8 to 17077] | 15355.8 [13623.7 to 19755.8] | 13876.8 [9103 to 16381.2] | 14499.8 [11288.4 to 19325.6]
  NL63-RBD-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 61 | 10 | 44 | 77 | 97 | 20 | 23 | 19 | 55 | 33
  NL63-RBD-50-Y at Month 4-Total | 16049.2 [13916.5 to 20575.2] | 16792.5 [11795.5 to 20184.8] | 16101.2 [15348.4 to 17799.4] | 15638.1 [10814.6 to 18445.9] | 16153.2 [11497 to 19545] | 16189.5 [12415 to 19226] | 16206 [12923.2 to 18796] | 15900.2 [12352.1 to 18463.5] | 17928.2 [15974.5 to 20689.9] | 16009.5 [12006.6 to 18225.5] | 16867 [15559.8 to 20416.8]
  OC43-RBD-50-N at Month 0-Total: number analyzed (Participants) | 242 | 178 | 244 | 200 | 152 | 126 | 235 | 221 | 220 | 201 | 200
  OC43-RBD-50-N at Month 0-Total | 4186.9 [2478.1 to 6786.4] | 4099.1 [2372.1 to 6822.8] | 4223.5 [2477.2 to 6737.6] | 4186.9 [2459.5 to 6814.8] | 4116.1 [2459.5 to 6946.5] | 4630 [2549.4 to 7625.1] | 4232 [2482.1 to 6762] | 4132 [2480.5 to 6810.8] | 3974.1 [2340.8 to 6538.6] | 4412.8 [2502.5 to 6884.8] | 4099.1 [2339.8 to 6666.6]
  OC43-RBD-50-N at Month 2-Total: number analyzed (Participants) | 240 | 171 | 245 | 187 | 137 | 131 | 232 | 230 | 235 | 193 | 211
  OC43-RBD-50-N at Month 2-Total | 4366.9 [2376.6 to 7504.3] | 4089.5 [2295 to 7386.2] | 4240 [2375.2 to 7488.8] | 4196.2 [2393 to 7230.9] | 4069.5 [2286 to 7110.5] | 4187.5 [2291.9 to 7386.2] | 4389.8 [2388.2 to 7524.1] | 4231.5 [2290.5 to 7281.8] | 4187.5 [2295 to 7054.2] | 4086.2 [2279.8 to 7551] | 4086.2 [2282.9 to 7054.2]
  OC43-RBD-50-N at Month 4-Total: number analyzed (Participants) | 168 | 124 | 171 | 137 | 108 | 90 | 164 | 160 | 163 | 128 | 152
  OC43-RBD-50-N at Month 4-Total | 5278.5 [2654.6 to 8500.8] | 5197.2 [2654.6 to 8500.8] | 5084.2 [2647.1 to 8505.2] | 5180.8 [2734 to 8573] | 5197.2 [2716 to 8685.4] | 5014.6 [2362.6 to 7717.4] | 5172.2 [2760.1 to 8515.4] | 5074.1 [2289.9 to 7816.8] | 5068.2 [2428.5 to 7898.2] | 5076.2 [2234.1 to 7843.8] | 4994.2 [2261.9 to 7573.8]
  OC43-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 18 | 82 | 16 | 60 | 108 | 134 | 25 | 39 | 40 | 59 | 60
  OC43-RBD-50-Y at Month 0-Total | 2889 [1346.3 to 5184.4] | 4563.8 [2505.5 to 6532.6] | 2867.8 [2124.6 to 5668.1] | 3976.2 [2257.1 to 6190] | 4318.9 [2317.3 to 6505.1] | 3843 [2227.7 to 6062.1] | 3117.5 [1859.2 to 5219.5] | 4143.8 [2184 to 5491.8] | 4958 [2906.1 to 7416.4] | 3533.5 [1821.8 to 5099.1] | 4471.8 [2781.4 to 6984.4]
  OC43-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 19 | 88 | 14 | 72 | 122 | 128 | 27 | 29 | 24 | 66 | 48
  OC43-RBD-50-Y at Month 2-Total | 2733.8 [1846.8 to 6103.2] | 4774.8 [2637.4 to 7509.4] | 4265.9 [1875.8 to 7046.3] | 4748.1 [1748.1 to 7575.7] | 4790.9 [2488.2 to 7749.9] | 4374.5 [2389.3 to 7490.4] | 3227.8 [1492.9 to 6747.8] | 4783 [2449 to 8253.8] | 5511.6 [2727.1 to 8294.2] | 4810.8 [2777.8 to 6952.4] | 5194 [2882.6 to 8128.2]
  OC43-RBD-50-Y at Month 4-Total: number analyzed (Participants) | 13 | 57 | 10 | 44 | 73 | 91 | 17 | 21 | 18 | 53 | 29
  OC43-RBD-50-Y at Month 4-Total | 3639.8 [2210.8 to 4224.8] | 4980 [2560.2 to 7899.2] | 5997.9 [2683.6 to 7579.4] | 4952.2 [2275.2 to 7267.4] | 4980 [2296.8 to 7434] | 5359.5 [2804.6 to 8505.2] | 4119.2 [2193.2 to 7379.2] | 6604 [3837.5 to 10017.8] | 6917.4 [4145.6 to 9177.4] | 5267.5 [3179.2 to 10017.8] | 7069.8 [4119.2 to 10017.8]
  SARS-CoV-2 DB His-1000-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 346 | 268 | 204 | 188 | 328 | 324 | 324 | 280 | 293
  SARS-CoV-2 DB His-1000-N at Month 0-Total | 6112.2 [1395.9 to 18561.8] | 6626 [1401.4 to 18561.8] | 5654.9 [1394.4 to 18179.1] | 7577.5 [1538.4 to 20529.9] | 8402.5 [1684.8 to 20938.4] | 6269.5 [1204.9 to 19740.6] | 5736.8 [1261.7 to 18723.8] | 4846.8 [1054.8 to 17239.6] | 5605.8 [1207.1 to 18613.7] | 5408.8 [1307.9 to 17605.1] | 5630.5 [1183.2 to 19230.8]
  SARS-CoV-2 DB His-1000-N at Month 2-Total: number analyzed (Participants) | 256 | 184 | 261 | 200 | 150 | 136 | 247 | 240 | 248 | 204 | 224
  SARS-CoV-2 DB His-1000-N at Month 2-Total | 2192 [585.6 to 6499.6] | 2048.1 [584.8 to 6592.7] | 2039.8 [587.8 to 6414.5] | 2409.2 [609 to 8690.5] | 2440.4 [622.9 to 8932] | 1574.5 [365.7 to 6567.6] | 2033 [558.2 to 6439.5] | 1626.9 [410.2 to 5818.3] | 1742.2 [536.1 to 6508.9] | 1655.6 [536.1 to 6102.7] | 1712 [513.1 to 6729.4]
  SARS-CoV-2 DB His-1000-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 103 | 181 | 177 | 181 | 145 | 168
  SARS-CoV-2 DB His-1000-N at Month 4-Total | 969 [309.1 to 3808.6] | 1020.2 [323 to 3617.6] | 836.9 [283.9 to 3774.9] | 958.2 [313.6 to 4088.1] | 1157.8 [356.2 to 3716.5] | 796.8 [301.9 to 4101.5] | 969 [293.5 to 4083.2] | 691 [276.5 to 3621] | 870.5 [293.5 to 4100.2] | 764.8 [296.2 to 3814.2] | 845.4 [280.4 to 4100.9]
  SARS-CoV-2 DB His-1000-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 21 | 99 | 163 | 179 | 39 | 43 | 43 | 87 | 74
  SARS-CoV-2 DB His-1000-Y at Month 0-Total | 1174.4 [258.6 to 2923.2] | 4122.1 [1011.9 to 15666.8] | 390.8 [1 to 4847.5] | 2841.8 [506.4 to 10564.5] | 4012 [905.6 to 13077.2] | 4669.8 [1230.6 to 14181] | 3328.2 [690.5 to 9756.9] | 10169.5 [2653.2 to 21961.9] | 4199 [1002.8 to 12758] | 4847.5 [466.8 to 16765.2] | 4638.5 [1342.9 to 13059.7]
  SARS-CoV-2 DB His-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 91 | 14 | 75 | 125 | 139 | 28 | 35 | 27 | 71 | 51
  SARS-CoV-2 DB His-1000-Y at Month 2-Total | 588 [88.5 to 1688.6] | 1592.5 [436.8 to 5293.5] | 418.8 [100.9 to 907.6] | 1164.2 [360 to 3250.1] | 1388.8 [410.8 to 4213.2] | 2390.5 [608.2 to 5812.9] | 1520.5 [513.1 to 4649.2] | 2760.2 [1676.5 to 9347] | 1211.8 [475.2 to 4381.5] | 2616.8 [550.5 to 5819.9] | 2056.5 [613.8 to 4632.5]
  SARS-CoV-2 DB His-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 97 | 19 | 23 | 19 | 55 | 32
  SARS-CoV-2 DB His-1000-Y at Month 4-Total | 226.5 [133 to 663.2] | 648.9 [173.2 to 3811.4] | 595.2 [447.4 to 1263.6] | 517.9 [174.8 to 1819.3] | 648.9 [182.4 to 3541.8] | 870.5 [257.2 to 2800] | 638.5 [288.5 to 956.6] | 1931.5 [1077.5 to 6169.6] | 509.2 [264.1 to 1517.8] | 1160.8 [225.9 to 3445] | 789.4 [403.5 to 1675.4]
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 348 | 270 | 205 | 187 | 328 | 323 | 324 | 280 | 293
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 0-Total | 12799.8 [2044.1 to 22000] | 13604.2 [2192.4 to 22000] | 12849 [2153.2 to 22000] | 13088.5 [2391.6 to 22000] | 14063.8 [2494 to 22000] | 13531.5 [1927 to 22000] | 11886.9 [1883.5 to 22000] | 11614.5 [1806.4 to 22000] | 13518.9 [1948.5 to 22000] | 12524.4 [2102.8 to 22000] | 12249.8 [1882 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 2-Total: number analyzed (Participants) | 250 | 176 | 257 | 197 | 146 | 133 | 240 | 235 | 244 | 199 | 222
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 2-Total | 2712.6 [618.1 to 8031.9] | 3177.2 [690.5 to 8193.8] | 2496 [603.8 to 8006.8] | 2949.5 [664.2 to 7406.5] | 3634 [706.7 to 8431] | 2042.2 [534.8 to 6959.5] | 2276.8 [580.1 to 7335.4] | 2042.2 [527.4 to 6960.5] | 2578.4 [586.4 to 8015.1] | 2235.8 [570 to 6850.6] | 2188.6 [583.6 to 7803.4]
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 4-Total: number analyzed (Participants) | 177 | 130 | 180 | 148 | 115 | 98 | 172 | 168 | 172 | 140 | 159
  SARS-CoV-2 Nucleoprotein His-1000-N at Month 4-Total | 554 [238 to 2161] | 645.5 [290.6 to 2248.2] | 519.9 [236.1 to 2123.5] | 515.1 [262 to 2003] | 684.2 [291.4 to 2238.4] | 520.1 [238.6 to 2063.4] | 530.8 [237.7 to 1932.3] | 471.8 [209.9 to 1834.7] | 562.2 [237.1 to 2222.4] | 497.9 [235.9 to 2003] | 554 [236.1 to 2189.9]
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 19 | 97 | 162 | 180 | 39 | 44 | 43 | 87 | 74
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 0-Total | 2446.9 [257.4 to 14302.8] | 8591 [1481.6 to 22000] | 474.2 [176.1 to 4311.5] | 7330.2 [823 to 20153.2] | 8591 [1457.2 to 22000] | 11080.2 [1907.4 to 22000] | 11964.5 [2066.5 to 22000] | 18448.9 [3083.5 to 22000] | 5702.8 [1539.4 to 15439.5] | 10451.2 [448 to 22000] | 10848.6 [2425 to 22000]
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 12 | 72 | 123 | 136 | 29 | 34 | 25 | 70 | 47
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 2-Total | 743 [117.5 to 2214.2] | 1519 [420.2 to 5682.8] | 705.9 [181.1 to 2720.7] | 1769.8 [402.2 to 8091.2] | 1746.2 [431.5 to 5970.2] | 3119.4 [656.8 to 8048] | 3486.5 [671.8 to 8151.2] | 4889.4 [1580.3 to 9442.2] | 1078.5 [589.2 to 5049.2] | 2712.6 [678.6 to 9358.6] | 3296.5 [625.1 to 6635.5]
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 60 | 10 | 42 | 75 | 92 | 18 | 22 | 18 | 50 | 31
  SARS-CoV-2 Nucleoprotein His-1000-Y at Month 4-Total | 427.5 [190.8 to 617.2] | 409.4 [175.7 to 1094.6] | 506.2 [177.1 to 733.1] | 531.6 [106.3 to 1372.3] | 427.5 [169.4 to 1139.9] | 515.1 [229.3 to 1846.2] | 398.9 [200.6 to 2714.5] | 962.6 [497.5 to 4748.5] | 416.5 [190.1 to 881.5] | 573.9 [236.3 to 1794] | 442 [207.9 to 1308.5]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 0-Total: number analyzed (Participants) | 248 | 180 | 248 | 201 | 154 | 126 | 237 | 226 | 221 | 201 | 200
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 0-Total | 6729.6 [1411.3 to 17060.8] | 6397.5 [1429.2 to 17470.2] | 6116 [1474.4 to 16115.8] | 8441.2 [1513.8 to 18425] | 8630.4 [2155.9 to 18162.2] | 8091.1 [1719.6 to 18162.2] | 5885.8 [1262 to 17378.2] | 4892.4 [1014.9 to 15449.3] | 7081 [1383 to 17507.8] | 5452.5 [1233 to 16424] | 7897.2 [1411.3 to 17908.7]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 2-Total: number analyzed (Participants) | 257 | 183 | 263 | 201 | 150 | 136 | 246 | 240 | 249 | 204 | 225
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 2-Total | 2060.5 [555.5 to 6803] | 2018.8 [564.8 to 6822.1] | 2016 [553.9 to 6577.5] | 2361 [643.5 to 7825.2] | 2397.1 [681 to 8594.2] | 1742.1 [434.7 to 5788.2] | 2000 [474.8 to 6768.3] | 1595.6 [402.9 to 5788.2] | 1984 [489.8 to 6512.5] | 1653.2 [493.4 to 5788.2] | 1928.5 [489.5 to 7137.5]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 102 | 180 | 177 | 181 | 145 | 167
  SARS-CoV-2 S Hexapro_293F_PPF-1000-N at Month 4-Total | 948.5 [299.9 to 3899] | 1037.6 [319.8 to 3900.8] | 843.1 [273.7 to 3873.3] | 987.8 [317.9 to 4360.8] | 1192 [348.4 to 4310.1] | 828.2 [288.4 to 3829.6] | 889.8 [262.3 to 3975.6] | 636.2 [233.2 to 3523] | 852 [284.5 to 4194.8] | 651 [275 to 3667.2] | 834.2 [263.8 to 4296.1]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 0-Total: number analyzed (Participants) | 16 | 84 | 16 | 63 | 110 | 138 | 27 | 38 | 43 | 63 | 64
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 0-Total | 1027.9 [84.6 to 2607.2] | 3242.9 [817.8 to 13852.2] | 278 [44.5 to 1890.9] | 2650.2 [577.4 to 7324] | 3143.1 [668.6 to 12575.8] | 3930.6 [829.8 to 12134.4] | 2550.5 [154.6 to 9876] | 6608.9 [2433 to 17724.8] | 2706 [632.1 to 8552] | 7081 [737.5 to 14116.5] | 2931.9 [739.4 to 9459.2]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 2-Total: number analyzed (Participants) | 18 | 92 | 12 | 74 | 125 | 139 | 29 | 35 | 26 | 71 | 50
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 2-Total | 464.8 [37.8 to 1475.5] | 1530.9 [387 to 4825.1] | 218.5 [76.9 to 846.8] | 857 [303.2 to 2440.4] | 1177.2 [385.2 to 4011] | 1984 [492.2 to 6733.6] | 1470.2 [509 to 3766.5] | 2944.5 [1505.6 to 10990.1] | 1153 [384.9 to 3760.7] | 2174 [479.8 to 7575.2] | 1835.5 [509.6 to 4802.1]
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 98 | 20 | 23 | 19 | 55 | 33
  SARS-CoV-2 S Hexapro_293F_PPF-1000-Y at Month 4-Total | 249 [128.5 to 426] | 435.4 [173.2 to 3385.9] | 351.6 [227.8 to 1244] | 329.8 [149.6 to 1633.1] | 369.9 [184.1 to 2818.1] | 688.2 [257.9 to 3793.9] | 459.1 [334.2 to 1232.5] | 2427 [483.6 to 8349.2] | 444.8 [240 to 1865] | 1209 [239.8 to 4150] | 636.2 [273.2 to 2592.5]
  SARS-CoV-2 S1 C His-1000-N at Month 0-Total: number analyzed (Participants) | 335 | 242 | 337 | 262 | 201 | 182 | 320 | 315 | 315 | 273 | 284
  SARS-CoV-2 S1 C His-1000-N at Month 0-Total | 5749.2 [1013.5 to 19426.4] | 5840.9 [1065.2 to 19804.8] | 5270.8 [1097.2 to 18916.2] | 6567 [1357.8 to 20734.9] | 7419.8 [1374.8 to 21077.8] | 4992 [934.4 to 19775.6] | 5146.4 [839.2 to 19649.8] | 4258.2 [704.8 to 17988] | 5061.5 [905.1 to 18752.1] | 4639.8 [992 to 18554.5] | 5023.5 [839.2 to 19084.6]
  SARS-CoV-2 S1 C His-1000-N at Month 2-Total: number analyzed (Participants) | 258 | 184 | 264 | 202 | 150 | 136 | 248 | 242 | 250 | 206 | 225
  SARS-CoV-2 S1 C His-1000-N at Month 2-Total | 1735.9 [351.6 to 6368.3] | 1719.5 [373.8 to 6311.1] | 1718.1 [347.8 to 6091.2] | 1913.9 [355.1 to 8352.1] | 2054.5 [414 to 8352.1] | 1464.6 [276.8 to 6040.8] | 1646.9 [318.8 to 6280.4] | 1455.4 [258.6 to 5586.8] | 1571.5 [302.7 to 6096.8] | 1464.6 [283 to 6096.8] | 1557.2 [286 to 6412.2]
  SARS-CoV-2 S1 C His-1000-N at Month 4-Total: number analyzed (Participants) | 187 | 138 | 190 | 156 | 122 | 103 | 181 | 177 | 181 | 145 | 168
  SARS-CoV-2 S1 C His-1000-N at Month 4-Total | 781 [232.8 to 4491] | 776.1 [259.2 to 4004.2] | 741.9 [210.4 to 4269.4] | 795.2 [240.6 to 4670.4] | 1001.6 [268.1 to 4269.4] | 718 [237.8 to 4642] | 775.5 [223.2 to 4568] | 597.2 [199.2 to 4099.2] | 752.2 [219.2 to 4647.5] | 683.2 [223.2 to 4116.8] | 741.9 [206.9 to 4670.4]
  SARS-CoV-2 S1 C His-1000-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 96 | 157 | 176 | 38 | 43 | 43 | 85 | 74
  SARS-CoV-2 S1 C His-1000-Y at Month 0-Total | 1047.2 [253.9 to 2268.5] | 3491.4 [665.9 to 15547.7] | 434.8 [22.2 to 2114.2] | 2149.2 [353.6 to 8389.4] | 3311.8 [563 to 11397] | 4395.6 [791.4 to 15229.9] | 3026.1 [618.1 to 7905.6] | 9263.5 [2702.5 to 22000] | 3529.5 [539.4 to 12927.5] | 7261 [525.8 to 17691.2] | 3837.6 [669.4 to 12453.1]
  SARS-CoV-2 S1 C His-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 13 | 75 | 127 | 141 | 29 | 35 | 27 | 71 | 52
  SARS-CoV-2 S1 C His-1000-Y at Month 2-Total | 324 [66.5 to 1153.2] | 1460.2 [236.8 to 5483.8] | 175.8 [87 to 776.5] | 776.5 [205.4 to 2233.6] | 995.8 [220.2 to 4688.8] | 1748.8 [324 to 5654.2] | 979.5 [268.5 to 4179.8] | 4179.8 [1485.5 to 11767.1] | 1180.2 [274.2 to 5120.1] | 2153.2 [439.2 to 5506.8] | 1527 [318.6 to 5453.1]
  SARS-CoV-2 S1 C His-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 62 | 10 | 44 | 78 | 97 | 19 | 23 | 19 | 55 | 32
  SARS-CoV-2 S1 C His-1000-Y at Month 4-Total | 223.2 [126.8 to 573] | 502.9 [135.1 to 4529.5] | 404.5 [287.8 to 1558.1] | 400.1 [113 to 1795.1] | 429 [135.1 to 3779.6] | 771.2 [191 to 3485.8] | 392 [195.5 to 950.2] | 1766.5 [703.8 to 8320.6] | 425.2 [202.1 to 1531.5] | 1073 [161.1 to 4140.2] | 607.5 [232.6 to 1822.1]
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 0-Total: number analyzed (Participants) | 341 | 245 | 345 | 267 | 203 | 187 | 327 | 322 | 322 | 278 | 291
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 0-Total | 6277.8 [1428.5 to 15321.2] | 5957.2 [1353.8 to 14702] | 5957.2 [1476.2 to 14716.8] | 6797.8 [1605.9 to 16543.5] | 6667.5 [1605.9 to 15640.6] | 5303.8 [1316 to 15341.2] | 5731 [1194.5 to 15326] | 5030.1 [984.8 to 14531.9] | 5896.4 [1303.1 to 15346.5] | 4911.9 [1297.1 to 14660.5] | 5892.2 [1282.2 to 15384.6]
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 2-Total: number analyzed (Participants) | 249 | 177 | 255 | 197 | 146 | 130 | 238 | 230 | 242 | 194 | 219
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 2-Total | 2590 [656.5 to 8193.8] | 2470 [656.5 to 8218.5] | 2552.8 [595.2 to 8034.6] | 2753.5 [555.2 to 9210] | 2573.2 [697.2 to 9068.9] | 1726.5 [505.6 to 8188] | 2510.6 [544.8 to 8164.3] | 2272.1 [414.4 to 7757.5] | 2573.2 [573.6 to 8164.3] | 1912.4 [544.8 to 7761.7] | 2470 [548.2 to 8157.9]
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 4-Total: number analyzed (Participants) | 176 | 129 | 178 | 146 | 114 | 95 | 170 | 165 | 170 | 136 | 158
  SARS-CoV-2 S1S2 ECD His-1000-N at Month 4-Total | 1046.5 [277.2 to 4434.6] | 1147 [359.3 to 4412] | 945.4 [246.9 to 4309.5] | 1046.5 [329.3 to 4479.9] | 1148.8 [360 to 4479.9] | 884.8 [312.2 to 4401.8] | 945.4 [214.2 to 4406.9] | 884.8 [185.2 to 4132.5] | 1004.9 [261.8 to 4816.6] | 876 [277.2 to 4271.5] | 945.4 [261.8 to 4406.9]
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 20 | 98 | 162 | 178 | 38 | 43 | 43 | 87 | 74
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 0-Total | 1058.1 [230.9 to 3826] | 4785.8 [790.2 to 14319.4] | 340.1 [27.9 to 4403.9] | 3834.1 [392.4 to 10674.8] | 4569.5 [642.3 to 12663.8] | 5896.4 [914.8 to 13916] | 5444.2 [1243.5 to 10841.9] | 9464 [3187.6 to 16543.5] | 3761 [535.5 to 10641.1] | 7128.5 [834.1 to 13892.2] | 5030.1 [677.1 to 12021.8]
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 2-Total: number analyzed (Participants) | 16 | 88 | 10 | 68 | 119 | 135 | 27 | 35 | 23 | 71 | 46
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 2-Total | 517.6 [148.9 to 2100.6] | 2524.2 [321.5 to 7310] | 411.1 [258.9 to 5514.1] | 1542 [565 to 3908.2] | 1917.5 [439.4 to 6580.4] | 2753.5 [626.8 to 7757.4] | 2286 [646.5 to 7051.5] | 2875 [1687.5 to 13120.5] | 1364.5 [305.6 to 3685.8] | 3353.2 [585.1 to 8034.6] | 2411.6 [611.9 to 6926.1]
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 4-Total: number analyzed (Participants) | 12 | 59 | 10 | 42 | 74 | 93 | 18 | 23 | 18 | 52 | 30
  SARS-CoV-2 S1S2 ECD His-1000-Y at Month 4-Total | 292.5 [64.6 to 506.6] | 573.5 [151.6 to 4182] | 479.5 [132.8 to 4063.2] | 577.6 [137.1 to 2494.4] | 619.4 [161.2 to 4130.2] | 985.8 [170.2 to 4123.5] | 707.4 [336.4 to 2884.1] | 1651 [683.1 to 6957.1] | 685.2 [162 to 1241.5] | 1212.5 [165.2 to 4377.2] | 893.4 [173.6 to 3046.6]
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 0-Total: number analyzed (Participants) | 345 | 249 | 349 | 271 | 207 | 187 | 330 | 324 | 326 | 282 | 295
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 0-Total | 14710.5 [5851 to 22000] | 14693.8 [5594.5 to 22000] | 14647.8 [6049.2 to 22000] | 17197.8 [6452.1 to 22000] | 17197.8 [6562 to 22000] | 12621.5 [5571.5 to 22000] | 14620.6 [5322.3 to 22000] | 12577.9 [4422.8 to 22000] | 14418.5 [5569.6 to 22000] | 12974.4 [5580.1 to 22000] | 13901.5 [5169.9 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 2-Total: number analyzed (Participants) | 258 | 184 | 264 | 202 | 151 | 137 | 248 | 242 | 251 | 205 | 227
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 2-Total | 8793 [2807.7 to 19804.5] | 8316.5 [3213.8 to 19446.9] | 8364.6 [2783.6 to 18903.7] | 8985.2 [2959.4 to 21977.7] | 9365.2 [3355.8 to 21955.4] | 7229 [2497.5 to 18788.5] | 8293.9 [2528.4 to 18809.6] | 7503.6 [2407.3 to 18640.9] | 8299.5 [2596.5 to 19108.4] | 7492.8 [2497.5 to 18579.2] | 7791 [2559.6 to 18934.6]
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 4-Total: number analyzed (Participants) | 189 | 139 | 192 | 158 | 123 | 103 | 182 | 178 | 183 | 146 | 169
  SARS-CoV-2 spike (PreS Nexelis)-1000-N at Month 4-Total | 4139.5 [1453.5 to 12774] | 4330.5 [1577.2 to 12902.2] | 3959.6 [1368.2 to 12176.1] | 4351 [1561.1 to 13770.2] | 5145 [1720.5 to 13932.6] | 3484 [1391.1 to 12454.6] | 3991.9 [1217 to 12655.1] | 3081.1 [1132.3 to 11488] | 3935.8 [1391.1 to 13703.2] | 3145.1 [1389.2 to 11574.7] | 3495.2 [1311 to 13569.2]
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 20 | 98 | 162 | 182 | 39 | 45 | 43 | 87 | 74
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 0-Total | 4467.4 [1171 to 9711.5] | 11566.1 [3761.4 to 22000] | 1821.1 [250.3 to 6792.7] | 9321.1 [1993.9 to 19944.7] | 10636 [3449.1 to 22000] | 14039.4 [4790.8 to 22000] | 11599 [4053.8 to 19094.5] | 19488.8 [9478.8 to 22000] | 12534.2 [4142.6 to 22000] | 15897.5 [3136.4 to 22000] | 14175.8 [5279.6 to 22000]
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 93 | 13 | 75 | 126 | 140 | 29 | 35 | 26 | 72 | 50
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 2-Total | 2182.5 [189 to 5763.9] | 7004 [1692.2 to 17791] | 1718.8 [240.5 to 5993.8] | 5330.8 [2061 to 12400.8] | 5994.6 [2407.3 to 14209] | 8793 [3058.1 to 18745.2] | 7004 [2798.8 to 16619.2] | 11160.5 [6801.9 to 20498.2] | 5687 [1814.8 to 14112.8] | 9950.8 [3375.2 to 19247.2] | 8293.9 [2418.6 to 17063.8]
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 99 | 20 | 24 | 19 | 56 | 33
  SARS-CoV-2 spike (PreS Nexelis)-1000-Y at Month 4-Total | 1020 [300.2 to 2101.5] | 2475.5 [654.2 to 11270.1] | 1830 [852.5 to 6023.1] | 2116.6 [698 to 7486.7] | 2238.8 [737.1 to 10305] | 3983.5 [1111 to 11925] | 2599.9 [1850.8 to 6494.4] | 7803.8 [2931.2 to 18528] | 2206.5 [1100.2 to 5812.5] | 5903.2 [920.6 to 13074.4] | 3783 [1289 to 9704]
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 0-Total: number analyzed (Participants) | 251 | 182 | 252 | 205 | 156 | 128 | 240 | 231 | 225 | 204 | 203
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 0-Total | 5490.5 [841 to 22000] | 5184.6 [757.2 to 22000] | 5305.8 [868.9 to 22000] | 6094.2 [996.5 to 22000] | 7176 [1151.7 to 22000] | 7429.1 [1142.4 to 22000] | 5216.2 [863.4 to 22000] | 4557 [502.2 to 21406] | 5490.5 [868 to 22000] | 5190.6 [823.8 to 22000] | 5783 [858.8 to 22000]
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 2-Total: number analyzed (Participants) | 250 | 177 | 257 | 198 | 146 | 132 | 241 | 234 | 242 | 201 | 220
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 2-Total | 1003.4 [103.7 to 5128] | 986.2 [100.8 to 4982.8] | 986.2 [101 to 4982.8] | 1344 [108.4 to 7489.8] | 1396.9 [103.7 to 7881.1] | 793.2 [90.9 to 6866.3] | 986.2 [101 to 4494.8] | 665.9 [68.8 to 4359.7] | 1003.4 [93.4 to 5128] | 805.5 [92.2 to 5145] | 979 [90.9 to 5178.8]
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 4-Total: number analyzed (Participants) | 188 | 138 | 191 | 157 | 122 | 103 | 181 | 178 | 182 | 146 | 168
  SARS-CoV-2-NTD-AVI Biotin-1000-N at Month 4-Total | 338.8 [38.4 to 2167.5] | 368.2 [52.4 to 2176.9] | 324 [32.4 to 2174.8] | 371.5 [46 to 2540.2] | 383.6 [59.6 to 2585.6] | 379.2 [50.9 to 2174.8] | 371.5 [38.2 to 2189.2] | 258.8 [22.1 to 1965.8] | 358.5 [29.4 to 2155.2] | 299.4 [38.9 to 2087.9] | 328 [26 to 2167.5]
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 0-Total: number analyzed (Participants) | 17 | 86 | 16 | 63 | 112 | 140 | 28 | 37 | 43 | 64 | 65
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 0-Total | 245.8 [3 to 1931] | 4697.5 [394.7 to 20450.7] | 173 [8.7 to 1331.1] | 1493.2 [175.9 to 8039.2] | 3231.6 [244.4 to 15086] | 3469.6 [329.1 to 17448.8] | 1559.1 [46.1 to 8833.2] | 8441 [1834 to 22000] | 2025.2 [187.2 to 10074.1] | 4045.6 [274.6 to 18452.3] | 2676.8 [375 to 11769.2]
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 2-Total: number analyzed (Participants) | 19 | 92 | 12 | 71 | 123 | 137 | 28 | 35 | 27 | 68 | 49
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 2-Total | 92.2 [3.4 to 715.9] | 692.4 [43.6 to 3752.1] | 39 [9.6 to 334.1] | 355 [24.1 to 1465.6] | 454.2 [55.1 to 2194.9] | 883.8 [101 to 4256] | 313.1 [18.1 to 3626.2] | 1859.5 [827.4 to 9648.6] | 361.2 [67.8 to 3031.5] | 1046 [88.1 to 3826.2] | 437.2 [163.5 to 3292.5]
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 4-Total: number analyzed (Participants) | 13 | 63 | 10 | 44 | 79 | 98 | 20 | 23 | 19 | 55 | 33
  SARS-CoV-2-NTD-AVI Biotin-1000-Y at Month 4-Total | 21.2 [2.5 to 377.2] | 252.5 [19.5 to 1865] | 172.6 [12.6 to 523.1] | 171 [6 to 601.3] | 189.2 [19.5 to 1354.6] | 275.8 [18.8 to 1964.2] | 99.8 [16.8 to 456.2] | 1242 [256.1 to 4546.8] | 152.8 [31.8 to 387.8] | 324 [4 to 2069.9] | 259.8 [40 to 1770.5]

48. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgG3) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
Participants
  2019-nCoV S/293F-50-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 175 | 166 | 123 | 112 | 166 | 157 | 160 | 150 | 153
  2019-nCoV S/293F-50-N at Month 0-Peru | 160 | 119 | 165 | 157 | 118 | 107 | 157 | 147 | 150 | 144 | 143
  2019-nCoV S/293F-50-N at Month 0-Total: number analyzed (Participants) | 345 | 249 | 348 | 271 | 206 | 187 | 330 | 323 | 326 | 282 | 296
  2019-nCoV S/293F-50-N at Month 0-Total | 312 | 225 | 316 | 248 | 191 | 172 | 295 | 288 | 290 | 262 | 263
  2019-nCoV S/293F-50-N at Month 0-USA: number analyzed (Participants) | 176 | 125 | 173 | 105 | 83 | 75 | 164 | 166 | 166 | 132 | 143
  2019-nCoV S/293F-50-N at Month 0-USA | 152 | 106 | 151 | 91 | 73 | 65 | 138 | 141 | 140 | 118 | 120
  2019-nCoV S/293F-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  2019-nCoV S/293F-50-N at Month 2-Peru | 24 | 20 | 26 | 24 | 19 | 18 | 26 | 22 | 24 | 23 | 23
  2019-nCoV S/293F-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  2019-nCoV S/293F-50-N at Month 2-Total | 78 | 61 | 77 | 51 | 41 | 46 | 74 | 74 | 76 | 62 | 70
  2019-nCoV S/293F-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  2019-nCoV S/293F-50-N at Month 2-USA | 54 | 41 | 51 | 27 | 22 | 28 | 48 | 52 | 52 | 39 | 47
  2019-nCoV S/293F-50-Y at Month 0-Peru: number analyzed (Participants) | 6 | 51 | 0 | 9 | 52 | 63 | 9 | 18 | 15 | 25 | 22
  2019-nCoV S/293F-50-Y at Month 0-Peru | 5 | 46 | 0 | 8 | 47 | 58 | 8 | 18 | 15 | 21 | 22
  2019-nCoV S/293F-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 21 | 98 | 163 | 182 | 39 | 46 | 43 | 87 | 73
  2019-nCoV S/293F-50-Y at Month 0-Total | 18 | 105 | 14 | 82 | 139 | 158 | 35 | 42 | 40 | 68 | 67
  2019-nCoV S/293F-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  2019-nCoV S/293F-50-Y at Month 0-USA | 13 | 59 | 14 | 74 | 92 | 100 | 27 | 24 | 25 | 47 | 45
  2019-nCoV S/293F-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  2019-nCoV S/293F-50-Y at Month 2-Peru | 2 | 6 | 0 | 2 | 7 | 8 | 0 | 4 | 2 | 3 | 3
  2019-nCoV S/293F-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  2019-nCoV S/293F-50-Y at Month 2-Total | 5 | 22 | 6 | 32 | 42 | 37 | 9 | 9 | 7 | 21 | 13
  2019-nCoV S/293F-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  2019-nCoV S/293F-50-Y at Month 2-USA | 3 | 16 | 6 | 30 | 35 | 29 | 9 | 5 | 5 | 18 | 10
  SARS-CoV-2 DB His-50-N at Month 0-Peru: number analyzed (Participants) | 168 | 123 | 175 | 166 | 122 | 112 | 166 | 158 | 160 | 150 | 152
  SARS-CoV-2 DB His-50-N at Month 0-Peru | 148 | 109 | 154 | 147 | 108 | 98 | 146 | 137 | 139 | 135 | 131
  SARS-CoV-2 DB His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 248 | 348 | 271 | 205 | 187 | 330 | 324 | 326 | 282 | 295
  SARS-CoV-2 DB His-50-N at Month 0-Total | 279 | 199 | 283 | 226 | 170 | 150 | 266 | 255 | 258 | 232 | 231
  SARS-CoV-2 DB His-50-N at Month 0-USA: number analyzed (Participants) | 176 | 125 | 173 | 105 | 83 | 75 | 164 | 166 | 166 | 132 | 143
  SARS-CoV-2 DB His-50-N at Month 0-USA | 131 | 90 | 129 | 79 | 62 | 52 | 120 | 118 | 119 | 97 | 100
  SARS-CoV-2 DB His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 DB His-50-N at Month 2-Peru | 14 | 11 | 14 | 12 | 10 | 9 | 14 | 12 | 12 | 11 | 12
  SARS-CoV-2 DB His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 DB His-50-N at Month 2-Total | 43 | 33 | 42 | 28 | 23 | 20 | 39 | 39 | 40 | 32 | 35
  SARS-CoV-2 DB His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 DB His-50-N at Month 2-USA | 29 | 22 | 28 | 16 | 13 | 11 | 25 | 27 | 28 | 21 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 17 | 15 | 25 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Peru | 6 | 45 | 0 | 7 | 46 | 56 | 8 | 17 | 15 | 19 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 182 | 39 | 45 | 43 | 87 | 74
  SARS-CoV-2 DB His-50-Y at Month 0-Total | 16 | 96 | 12 | 69 | 125 | 145 | 29 | 40 | 37 | 63 | 64
  SARS-CoV-2 DB His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 DB His-50-Y at Month 0-USA | 10 | 51 | 12 | 62 | 79 | 89 | 21 | 23 | 22 | 44 | 41
  SARS-CoV-2 DB His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 DB His-50-Y at Month 2-Peru | 0 | 3 | 0 | 2 | 4 | 5 | 0 | 2 | 2 | 3 | 2
  SARS-CoV-2 DB His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 DB His-50-Y at Month 2-Total | 2 | 12 | 3 | 17 | 22 | 25 | 6 | 6 | 5 | 13 | 10
  SARS-CoV-2 DB His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 DB His-50-Y at Month 2-USA | 2 | 9 | 3 | 15 | 18 | 20 | 6 | 4 | 3 | 10 | 8
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru: number analyzed (Participants) | 169 | 125 | 176 | 167 | 124 | 113 | 167 | 159 | 161 | 152 | 153
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru | 160 | 120 | 166 | 158 | 119 | 109 | 158 | 149 | 151 | 147 | 143
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 249 | 348 | 271 | 206 | 187 | 330 | 324 | 326 | 283 | 295
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total | 316 | 231 | 319 | 251 | 194 | 176 | 301 | 293 | 295 | 267 | 267
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA: number analyzed (Participants) | 175 | 124 | 172 | 104 | 82 | 74 | 163 | 165 | 165 | 131 | 142
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA | 156 | 111 | 153 | 93 | 75 | 67 | 143 | 144 | 144 | 120 | 124
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru | 20 | 16 | 22 | 20 | 15 | 14 | 22 | 18 | 20 | 19 | 19
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total | 72 | 57 | 71 | 46 | 37 | 41 | 68 | 67 | 70 | 55 | 65
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA | 52 | 41 | 49 | 26 | 22 | 27 | 46 | 49 | 50 | 36 | 46
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 63 | 9 | 17 | 15 | 24 | 23
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru | 6 | 46 | 0 | 8 | 47 | 57 | 8 | 17 | 15 | 19 | 23
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 182 | 39 | 45 | 43 | 86 | 74
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total | 19 | 104 | 16 | 84 | 141 | 159 | 34 | 42 | 40 | 68 | 68
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA | 13 | 58 | 16 | 76 | 94 | 102 | 26 | 25 | 25 | 49 | 45
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru | 2 | 6 | 0 | 2 | 7 | 8 | 0 | 4 | 2 | 3 | 3
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total | 4 | 19 | 5 | 30 | 39 | 35 | 8 | 9 | 6 | 21 | 11
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA | 2 | 13 | 5 | 28 | 32 | 27 | 8 | 5 | 4 | 18 | 8
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru: number analyzed (Participants) | 167 | 123 | 174 | 165 | 122 | 112 | 165 | 158 | 159 | 150 | 151
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru | 152 | 114 | 158 | 151 | 113 | 103 | 151 | 142 | 143 | 139 | 135
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total: number analyzed (Participants) | 342 | 247 | 346 | 269 | 204 | 187 | 328 | 324 | 324 | 282 | 293
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total | 287 | 207 | 290 | 232 | 177 | 158 | 274 | 265 | 265 | 240 | 237
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA: number analyzed (Participants) | 175 | 124 | 172 | 104 | 82 | 75 | 163 | 166 | 165 | 132 | 142
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA | 135 | 93 | 132 | 81 | 64 | 55 | 123 | 123 | 122 | 101 | 102
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru | 18 | 14 | 18 | 16 | 13 | 13 | 18 | 16 | 16 | 15 | 16
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total | 54 | 41 | 54 | 37 | 29 | 29 | 49 | 50 | 52 | 42 | 47
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA | 36 | 27 | 36 | 21 | 16 | 16 | 31 | 34 | 36 | 27 | 31
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 62 | 9 | 16 | 15 | 24 | 23
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru | 6 | 44 | 0 | 7 | 45 | 55 | 7 | 16 | 15 | 19 | 23
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 180 | 39 | 43 | 43 | 85 | 74
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total | 16 | 96 | 13 | 71 | 126 | 145 | 29 | 38 | 38 | 63 | 66
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 118 | 30 | 27 | 28 | 61 | 51
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA | 10 | 52 | 13 | 64 | 81 | 90 | 22 | 22 | 23 | 44 | 43
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru | 0 | 4 | 0 | 2 | 5 | 5 | 0 | 2 | 2 | 3 | 2
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total | 3 | 16 | 3 | 20 | 28 | 28 | 8 | 7 | 5 | 15 | 10
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA | 3 | 12 | 3 | 18 | 23 | 23 | 8 | 5 | 3 | 12 | 8
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru: number analyzed (Participants) | 170 | 125 | 177 | 168 | 124 | 113 | 168 | 159 | 162 | 152 | 154
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru | 153 | 114 | 159 | 152 | 113 | 101 | 151 | 141 | 144 | 139 | 136
  SARS-CoV-2 S1 C His-50-N at Month 0-Total: number analyzed (Participants) | 346 | 250 | 350 | 273 | 207 | 188 | 332 | 325 | 328 | 284 | 297
  SARS-CoV-2 S1 C His-50-N at Month 0-Total | 292 | 211 | 294 | 233 | 178 | 157 | 277 | 266 | 271 | 242 | 244
  SARS-CoV-2 S1 C His-50-N at Month 0-USA: number analyzed (Participants) | 176 | 125 | 173 | 105 | 83 | 75 | 164 | 166 | 166 | 132 | 143
  SARS-CoV-2 S1 C His-50-N at Month 0-USA | 139 | 97 | 135 | 81 | 65 | 56 | 126 | 125 | 127 | 103 | 108
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru | 18 | 14 | 19 | 17 | 13 | 12 | 19 | 15 | 17 | 16 | 17
  SARS-CoV-2 S1 C His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1 C His-50-N at Month 2-Total | 56 | 44 | 56 | 38 | 29 | 28 | 52 | 51 | 54 | 43 | 49
  SARS-CoV-2 S1 C His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S1 C His-50-N at Month 2-USA | 38 | 30 | 37 | 21 | 16 | 16 | 33 | 36 | 37 | 27 | 32
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru | 6 | 45 | 0 | 7 | 46 | 58 | 8 | 18 | 15 | 20 | 23
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 183 | 39 | 46 | 43 | 87 | 74
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total | 15 | 96 | 13 | 74 | 129 | 150 | 30 | 41 | 36 | 65 | 63
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA | 9 | 51 | 13 | 67 | 83 | 92 | 22 | 23 | 21 | 45 | 40
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru | 1 | 5 | 0 | 2 | 6 | 7 | 0 | 4 | 2 | 3 | 2
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total | 4 | 16 | 4 | 22 | 31 | 32 | 8 | 9 | 6 | 17 | 11
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA | 3 | 11 | 4 | 20 | 25 | 25 | 8 | 5 | 4 | 14 | 9
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru: number analyzed (Participants) | 170 | 125 | 177 | 168 | 124 | 113 | 168 | 159 | 162 | 152 | 154
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru | 159 | 117 | 165 | 157 | 116 | 107 | 157 | 147 | 150 | 145 | 142
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 348 | 271 | 205 | 186 | 329 | 322 | 326 | 281 | 295
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total | 314 | 226 | 317 | 249 | 190 | 171 | 296 | 291 | 293 | 263 | 263
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA: number analyzed (Participants) | 173 | 122 | 171 | 103 | 81 | 73 | 161 | 163 | 164 | 129 | 141
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA | 155 | 109 | 152 | 92 | 74 | 64 | 139 | 144 | 143 | 118 | 121
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru | 26 | 21 | 29 | 27 | 20 | 20 | 29 | 25 | 27 | 25 | 26
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total | 83 | 66 | 83 | 58 | 46 | 49 | 79 | 80 | 82 | 66 | 76
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA | 57 | 45 | 54 | 31 | 26 | 29 | 50 | 55 | 55 | 41 | 50
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru | 6 | 48 | 0 | 8 | 49 | 58 | 8 | 18 | 15 | 20 | 23
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 20 | 97 | 163 | 182 | 39 | 46 | 42 | 87 | 73
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total | 19 | 107 | 16 | 84 | 143 | 162 | 37 | 42 | 40 | 70 | 70
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 20 | 88 | 110 | 118 | 30 | 28 | 27 | 62 | 50
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA | 13 | 59 | 16 | 76 | 94 | 104 | 29 | 24 | 25 | 50 | 47
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru | 3 | 8 | 0 | 2 | 9 | 9 | 0 | 4 | 2 | 4 | 3
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total | 6 | 23 | 6 | 31 | 43 | 40 | 10 | 9 | 7 | 23 | 13
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA | 3 | 15 | 6 | 29 | 34 | 31 | 10 | 5 | 5 | 19 | 10
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru: number analyzed (Participants) | 170 | 125 | 177 | 168 | 124 | 113 | 168 | 159 | 162 | 152 | 154
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru | 161 | 120 | 167 | 159 | 119 | 108 | 159 | 149 | 152 | 146 | 144
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total: number analyzed (Participants) | 346 | 250 | 350 | 273 | 207 | 188 | 332 | 325 | 328 | 284 | 297
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total | 312 | 226 | 317 | 250 | 192 | 172 | 296 | 289 | 291 | 263 | 263
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA: number analyzed (Participants) | 176 | 125 | 173 | 105 | 83 | 75 | 164 | 166 | 166 | 132 | 143
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA | 151 | 106 | 150 | 91 | 73 | 64 | 137 | 140 | 139 | 117 | 119
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru | 23 | 19 | 25 | 23 | 18 | 16 | 25 | 21 | 23 | 21 | 22
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total | 75 | 58 | 74 | 49 | 39 | 42 | 71 | 71 | 73 | 58 | 67
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA | 52 | 39 | 49 | 26 | 21 | 26 | 46 | 50 | 50 | 37 | 45
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru | 6 | 47 | 0 | 8 | 48 | 59 | 8 | 18 | 15 | 21 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 183 | 39 | 46 | 43 | 87 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total | 19 | 105 | 14 | 81 | 139 | 159 | 35 | 42 | 40 | 68 | 68
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA | 13 | 58 | 14 | 73 | 91 | 100 | 27 | 24 | 25 | 47 | 45
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru | 2 | 6 | 0 | 2 | 7 | 9 | 0 | 4 | 2 | 4 | 3
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total | 5 | 22 | 6 | 31 | 41 | 38 | 9 | 9 | 7 | 22 | 13
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA | 3 | 16 | 6 | 29 | 34 | 29 | 9 | 5 | 5 | 18 | 10
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru: number analyzed (Participants) | 169 | 125 | 176 | 167 | 124 | 113 | 167 | 159 | 161 | 152 | 153
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru | 156 | 117 | 161 | 154 | 116 | 105 | 153 | 144 | 146 | 142 | 139
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total: number analyzed (Participants) | 345 | 250 | 349 | 272 | 207 | 188 | 331 | 325 | 327 | 284 | 296
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total | 297 | 215 | 297 | 237 | 182 | 164 | 279 | 272 | 275 | 248 | 249
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA: number analyzed (Participants) | 176 | 125 | 173 | 105 | 83 | 75 | 164 | 166 | 166 | 132 | 143
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA | 141 | 98 | 136 | 83 | 66 | 59 | 126 | 128 | 129 | 106 | 110
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru | 24 | 19 | 25 | 23 | 18 | 18 | 25 | 21 | 23 | 22 | 23
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total | 73 | 56 | 73 | 50 | 40 | 41 | 66 | 67 | 71 | 57 | 66
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA | 49 | 37 | 48 | 27 | 22 | 23 | 41 | 46 | 48 | 35 | 43
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 63 | 9 | 17 | 15 | 24 | 23
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru | 5 | 44 | 0 | 7 | 45 | 56 | 8 | 17 | 15 | 19 | 22
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 182 | 39 | 45 | 43 | 86 | 74
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total | 13 | 95 | 13 | 73 | 128 | 146 | 31 | 38 | 35 | 62 | 61
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 69 | 21 | 89 | 111 | 119 | 30 | 28 | 28 | 62 | 51
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA | 8 | 51 | 13 | 66 | 83 | 90 | 23 | 21 | 20 | 43 | 39
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru | 1 | 6 | 0 | 2 | 7 | 7 | 0 | 4 | 2 | 3 | 2
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total | 3 | 20 | 3 | 26 | 36 | 35 | 10 | 9 | 5 | 19 | 10
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA | 2 | 14 | 3 | 24 | 29 | 28 | 10 | 5 | 3 | 16 | 8

49. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgG3) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgG3) at Visit 1, 2, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
MFI
  2019-nCoV S/293F-50-N at Month 0-Total: number analyzed (Participants) | 345 | 249 | 348 | 271 | 206 | 187 | 330 | 323 | 326 | 282 | 296
  2019-nCoV S/293F-50-N at Month 0-Total | 6714.8 [3175.5 to 12619.5] | 6505.5 [2988.5 to 11434] | 6657.1 [3173.7 to 12470.5] | 6717.8 [3218.6 to 12565.2] | 6796.4 [3091.3 to 11935.9] | 6335.5 [2958.2 to 12565.2] | 6576.2 [3091.3 to 12270] | 5847.5 [2812.1 to 11832.5] | 6703 [3085.7 to 12651] | 6254.2 [3177.9 to 11998.9] | 6703 [2948.6 to 12812.1]
  2019-nCoV S/293F-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  2019-nCoV S/293F-50-N at Month 2-Total | 3302.6 [1426.4 to 4901.2] | 3307 [1213.5 to 4617.2] | 3146.2 [1213.5 to 4824] | 3002.2 [595 to 4824] | 3240 [620.9 to 4776.5] | 2815.5 [1070.4 to 4376.5] | 3146.2 [1373 to 4673.1] | 3002.2 [726.6 to 4776.5] | 3193.1 [1311 to 4901.2] | 2880 [1040.9 to 4776.5] | 3074.2 [1246 to 4800.2]
  2019-nCoV S/293F-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 120 | 21 | 98 | 163 | 182 | 39 | 46 | 43 | 87 | 73
  2019-nCoV S/293F-50-Y at Month 0-Total | 5043.9 [1256.1 to 6848] | 6335.1 [3284.1 to 13264.6] | 3630 [320.5 to 7354.2] | 5487.2 [2629.2 to 11416.2] | 6175.8 [3056.6 to 12609.4] | 6524.4 [3232.5 to 11935.9] | 5381.5 [2736.1 to 12524.9] | 9506.1 [5069.1 to 16105.3] | 5317.5 [3193.5 to 8108.1] | 6800 [2082.1 to 12771] | 5585.5 [3350.2 to 9871.2]
  2019-nCoV S/293F-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  2019-nCoV S/293F-50-Y at Month 2-Total | 983.1 [1 to 2103.1] | 2880 [1377.8 to 5805.1] | 3467.5 [1951 to 3837.9] | 3467.5 [1718.5 to 4519.4] | 3079.8 [1447.8 to 4617.2] | 3467.5 [1343.5 to 6583.5] | 3472.5 [429.8 to 5169.8] | 3838.8 [3079.8 to 4617.2] | 3273.6 [1220.7 to 3636.6] | 3562 [1447.8 to 4617.2] | 3327.5 [1628.5 to 3954.7]
  229E-RBD-50-N at Month 0-Total: number analyzed (Participants) | 335 | 242 | 338 | 264 | 199 | 184 | 322 | 314 | 317 | 276 | 288
  229E-RBD-50-N at Month 0-Total | 250.5 [39.1 to 489.1] | 252.1 [44.6 to 473.3] | 251.5 [36 to 510.5] | 246.4 [35.2 to 473.1] | 251.2 [43.2 to 453] | 252.9 [60.1 to 440.6] | 252.1 [40 to 482.2] | 224.2 [34.6 to 460.2] | 225 [31.5 to 471.2] | 241.4 [60.1 to 459.6] | 233.8 [37 to 471.6]
  229E-RBD-50-N at Month 2-Total: number analyzed (Participants) | 91 | 73 | 92 | 65 | 51 | 54 | 86 | 90 | 91 | 74 | 85
  229E-RBD-50-N at Month 2-Total | 1 [1 to 24.1] | 1 [1 to 19.8] | 1 [1 to 19.8] | 1 [1 to 6] | 1 [1 to 11.4] | 1 [1 to 1] | 1 [1 to 19] | 1 [1 to 26.3] | 1 [1 to 18.2] | 1 [1 to 26.3] | 1 [1 to 1]
  229E-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 20 | 94 | 159 | 174 | 36 | 44 | 41 | 82 | 70
  229E-RBD-50-Y at Month 0-Total | 116.5 [1 to 501.5] | 200.2 [4.8 to 521.3] | 160.9 [35.9 to 306.8] | 220.6 [45.9 to 536.4] | 221 [19.2 to 548] | 220.6 [4.6 to 576.2] | 192.1 [24.3 to 724.8] | 333 [70.5 to 637.6] | 345.2 [109.5 to 633.5] | 202.4 [1 to 599.9] | 293 [33.6 to 574.2]
  229E-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 26 | 7 | 34 | 48 | 45 | 13 | 9 | 8 | 25 | 14
  229E-RBD-50-Y at Month 2-Total | 1 [1 to 1] | 1 [1 to 15.1] | 1 [1 to 33] | 1 [1 to 60.5] | 1 [1 to 51.5] | 1 [1 to 160.5] | 1 [1 to 19.8] | 1 [1 to 1] | 1 [1 to 31.1] | 1 [1 to 16.8] | 10.4 [1 to 358.9]
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 248 | 348 | 271 | 205 | 188 | 330 | 323 | 326 | 283 | 296
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total | 13.8 [1 to 100.4] | 17.2 [1 to 80.3] | 12.1 [1 to 100.4] | 2.5 [1 to 75.9] | 4.2 [1 to 72.2] | 23.4 [1 to 108.6] | 13.8 [1 to 99.6] | 13.8 [1 to 102.1] | 9.9 [1 to 96.2] | 21.2 [1 to 102.1] | 12.1 [1 to 104.1]
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 181 | 39 | 46 | 43 | 86 | 73
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total | 1 [1 to 59] | 1 [1 to 116.8] | 1 [1 to 59] | 24 [1 to 150.2] | 18.1 [1 to 133.3] | 1 [1 to 73.2] | 1 [1 to 101.1] | 1 [1 to 70.3] | 26 [1 to 113.4] | 1 [1 to 67.9] | 5.2 [1 to 77.8]
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1042.5] | 1 [1 to 33.5] | 1 [1 to 1] | 1 [1 to 31.2] | 1 [1 to 1] | 1 [1 to 1] | 15.2 [1 to 148.9] | 1 [1 to 209.5] | 1 [1 to 35.9]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 342 | 247 | 346 | 270 | 204 | 187 | 329 | 321 | 324 | 283 | 295
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total | 389.4 [132.7 to 1182] | 396.8 [145.5 to 973.8] | 370.1 [129.1 to 1109.1] | 341.9 [114.4 to 947.2] | 359 [141.6 to 939.8] | 419.2 [157.8 to 1087.6] | 369 [141.8 to 1088.2] | 369 [127.8 to 1028.8] | 376.9 [126.9 to 1125.8] | 395.8 [148.2 to 1206.4] | 377.5 [137.5 to 1121.6]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total | 167.4 [1 to 826.1] | 186.8 [1 to 584] | 156.2 [1 to 652.8] | 115.2 [1 to 479.8] | 161.5 [1 to 532.5] | 192.5 [1 to 793.2] | 164.5 [1 to 835.1] | 186.8 [1 to 848.9] | 160.9 [1 to 673.4] | 161.5 [1 to 694.1] | 158.2 [1 to 714.8]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 97 | 163 | 180 | 38 | 46 | 43 | 84 | 72
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total | 312 [125.5 to 707.8] | 349.4 [102.9 to 1831.8] | 514.2 [147.2 to 1809] | 450.2 [177.5 to 2485.8] | 432.2 [121.8 to 1854.6] | 337.4 [89.4 to 1169.6] | 478.1 [44.3 to 1963.3] | 490.9 [167.3 to 1806.4] | 371.2 [204.8 to 1259.9] | 354.2 [92 to 982.8] | 354.4 [125.2 to 1194.7]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total | 1 [1 to 541.8] | 112.2 [1 to 1257.8] | 1346.5 [326.8 to 1859.5] | 371 [60.6 to 1827.6] | 164.5 [1 to 1255.8] | 150 [1 to 819.2] | 150 [1 to 502.8] | 63 [1 to 150] | 651.2 [140.6 to 1392.9] | 170.2 [35.8 to 1532.2] | 293.4 [121.7 to 1214.7]
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 248 | 348 | 271 | 205 | 188 | 330 | 323 | 326 | 283 | 296
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total | 1 [1 to 53.9] | 1 [1 to 54.2] | 1 [1 to 51.7] | 1 [1 to 42.1] | 1 [1 to 41.5] | 1 [1 to 64.6] | 1 [1 to 52.1] | 1 [1 to 54.2] | 1 [1 to 50.4] | 1 [1 to 58.5] | 1 [1 to 52.4]
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 181 | 39 | 46 | 43 | 86 | 73
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total | 1 [1 to 15.8] | 1 [1 to 44.5] | 4.5 [1 to 75.5] | 7.1 [1 to 76.8] | 1 [1 to 58.4] | 1 [1 to 35.5] | 1 [1 to 51.4] | 1 [1 to 11.5] | 14 [1 to 57] | 1 [1 to 22.8] | 1 [1 to 51.5]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 360.4] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 76.1] | 1 [1 to 14.8] | 1 [1 to 193.7]
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 343 | 248 | 347 | 271 | 205 | 187 | 330 | 322 | 325 | 283 | 295
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total | 519.8 [124.5 to 1842.5] | 480.6 [131.5 to 1640.4] | 476 [124.5 to 1752.2] | 410.8 [93.9 to 1394.8] | 419.5 [118.5 to 1479] | 475.8 [164.2 to 1686.9] | 492.1 [128.3 to 1757.1] | 480.6 [131.9 to 1715.2] | 448.5 [113.2 to 1882.8] | 500.8 [133.6 to 1791] | 464.2 [117.6 to 1772.4]
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 91 | 72 | 92 | 64 | 50 | 54 | 85 | 89 | 91 | 74 | 85
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total | 12.2 [1 to 573.8] | 11.2 [1 to 571.9] | 2.9 [1 to 521.9] | 1 [1 to 352.9] | 5.6 [1 to 498.4] | 22.2 [1 to 575.6] | 10.2 [1 to 570] | 10.2 [1 to 577.5] | 1 [1 to 559.6] | 11.2 [1 to 564.8] | 1 [1 to 570]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 97 | 163 | 181 | 38 | 46 | 43 | 85 | 73
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total | 397.8 [105 to 1386.8] | 523.2 [94.3 to 2453.6] | 967 [105 to 2514.5] | 825.8 [272.2 to 4158.5] | 610.2 [127.4 to 3077.8] | 519.8 [93 to 1923.5] | 513.8 [12.1 to 2798.4] | 629.5 [65.6 to 3871.4] | 861.8 [224 to 1671.5] | 476 [98.2 to 1650.5] | 618.8 [131 to 1779.8]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 7 | 26 | 6 | 34 | 48 | 44 | 13 | 9 | 7 | 24 | 13
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total | 1 [1 to 172.9] | 2.9 [1 to 329.2] | 1326.5 [245.5 to 2615.1] | 233.1 [1 to 2884.8] | 8.5 [1 to 805.8] | 1 [1 to 457.8] | 1 [1 to 377.2] | 1 [1 to 222.5] | 222.5 [103 to 706.6] | 1 [1 to 683.3] | 222.5 [1 to 434.2]
  HKU1-RBD-50-N at Month 0-Total: number analyzed (Participants) | 339 | 246 | 341 | 267 | 204 | 182 | 323 | 316 | 320 | 276 | 290
  HKU1-RBD-50-N at Month 0-Total | 207 [59.1 to 384.9] | 207.4 [59.9 to 395.2] | 203.8 [46.2 to 380.5] | 203.8 [48.5 to 380.2] | 208.1 [59.4 to 380.1] | 207.1 [78.1 to 378.1] | 204 [45 to 372.1] | 191.6 [43.4 to 361.4] | 193 [39.9 to 374.4] | 205.1 [71.8 to 370.6] | 183.9 [40.4 to 387.1]
  HKU1-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HKU1-RBD-50-N at Month 2-Total | 1 [1 to 84.1] | 1 [1 to 55.8] | 1 [1 to 81.2] | 1 [1 to 68.8] | 1 [1 to 16.6] | 1 [1 to 1.6] | 1 [1 to 62.2] | 1 [1 to 75] | 1 [1 to 71.9] | 1 [1 to 75] | 1 [1 to 17.3]
  HKU1-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 95 | 158 | 180 | 39 | 46 | 42 | 86 | 72
  HKU1-RBD-50-Y at Month 0-Total | 123.5 [1 to 196.5] | 175.8 [18.7 to 356.3] | 150.5 [29.5 to 312.8] | 179.2 [31.6 to 385.1] | 177.5 [29.6 to 385.8] | 174 [13.2 to 411.1] | 167.2 [10 to 566.9] | 246.8 [1 to 569] | 213.4 [81.4 to 517.4] | 157.9 [1 to 445.2] | 212.2 [65.3 to 367.9]
  HKU1-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HKU1-RBD-50-Y at Month 2-Total | 1 [1 to 204.2] | 1 [1 to 107.9] | 1 [1 to 130.6] | 1 [1 to 129.8] | 1 [1 to 123] | 1 [1 to 233] | 1 [1 to 352] | 1 [1 to 123] | 1 [1 to 529.1] | 1 [1 to 123] | 62 [1 to 737.9]
  NL63-RBD-50-N at Month 0-Total: number analyzed (Participants) | 325 | 237 | 327 | 255 | 196 | 178 | 309 | 303 | 308 | 268 | 279
  NL63-RBD-50-N at Month 0-Total | 219.8 [21.8 to 447.5] | 224.5 [28.8 to 453] | 218.2 [17.8 to 448.2] | 200.8 [19.6 to 436.2] | 219.5 [20.7 to 447.1] | 208.9 [17.6 to 441.8] | 219.2 [17.5 to 444.8] | 214.8 [12.8 to 433] | 201.1 [11.8 to 433] | 202.6 [23.6 to 433] | 195.2 [11.6 to 433]
  NL63-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  NL63-RBD-50-N at Month 2-Total | 1 [1 to 62] | 1 [1 to 57.2] | 1 [1 to 57.2] | 1 [1 to 1] | 1 [1 to 6.1] | 1 [1 to 8] | 1 [1 to 30.1] | 1 [1 to 51.2] | 1 [1 to 48.2] | 1 [1 to 51.2] | 1 [1 to 8.7]
  NL63-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 21 | 109 | 19 | 91 | 150 | 168 | 37 | 43 | 38 | 78 | 67
  NL63-RBD-50-Y at Month 0-Total | 131.5 [1 to 245.5] | 193.2 [1 to 401.2] | 131.5 [1 to 381.2] | 258.2 [1 to 498.1] | 202.6 [1 to 427.6] | 217.2 [8.7 to 446.4] | 170 [1 to 514.2] | 245.5 [23.2 to 495.4] | 284.5 [32.3 to 548.6] | 246 [1 to 512.8] | 296.2 [20.4 to 534.6]
  NL63-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  NL63-RBD-50-Y at Month 2-Total | 1 [1 to 1] | 1 [1 to 8] | 1 [1 to 1] | 1 [1 to 131.6] | 1 [1 to 110.8] | 1 [1 to 110.8] | 1 [1 to 110.8] | 1 [1 to 1] | 1 [1 to 28.4] | 1 [1 to 11.2] | 1 [1 to 189.5]
  OC43-RBD-50-N at Month 0-Total: number analyzed (Participants) | 340 | 245 | 343 | 268 | 203 | 185 | 325 | 319 | 323 | 279 | 292
  OC43-RBD-50-N at Month 0-Total | 154.1 [1.2 to 358.6] | 152.2 [1.2 to 339.2] | 151.5 [1 to 361.1] | 150.6 [1 to 350.1] | 158.8 [3 to 337.5] | 158.8 [1 to 310.2] | 146.5 [1 to 339.2] | 142.8 [1 to 339.2] | 138.2 [1 to 323.6] | 156 [1.1 to 337.5] | 145.2 [1 to 323.6]
  OC43-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  OC43-RBD-50-N at Month 2-Total | 1 [1 to 21.4] | 1 [1 to 28.8] | 1 [1 to 16.8] | 1 [1 to 16.8] | 1 [1 to 22.8] | 1 [1 to 1] | 1 [1 to 7.2] | 1 [1 to 17.9] | 1 [1 to 17.3] | 1 [1 to 13.4] | 1 [1 to 1]
  OC43-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 96 | 161 | 179 | 39 | 45 | 41 | 85 | 72
  OC43-RBD-50-Y at Month 0-Total | 41.4 [1 to 237.8] | 123 [1 to 390.2] | 73.8 [1 to 233] | 136.6 [6.1 to 359.4] | 127 [1 to 380.8] | 130 [1 to 425.6] | 138.2 [1 to 476.8] | 159.8 [74 to 450.5] | 218.2 [22.8 to 520.8] | 121.5 [1 to 405.8] | 158.4 [1 to 464.4]
  OC43-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  OC43-RBD-50-Y at Month 2-Total | 1 [1 to 125.2] | 1 [1 to 1] | 10 [1 to 122.8] | 1 [1 to 33.8] | 1 [1 to 19] | 1 [1 to 121] | 1 [1 to 388] | 1 [1 to 48.5] | 5.5 [1 to 258.3] | 1 [1 to 48.5] | 29.5 [1 to 417.6]
  SARS-CoV-2 DB His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 248 | 348 | 271 | 205 | 187 | 330 | 324 | 326 | 282 | 295
  SARS-CoV-2 DB His-50-N at Month 0-Total | 1930 [666.7 to 4088.1] | 1917.8 [610.6 to 3822.1] | 1917.8 [666.7 to 4009.2] | 1963.8 [803.5 to 4047.9] | 2080 [803 to 4008.5] | 1815.5 [595.1 to 3818.5] | 1888.6 [654.5 to 3853.4] | 1757.4 [544.4 to 3732] | 1866.4 [550.7 to 3981.6] | 1859.2 [679.1 to 3786.4] | 1848.5 [534.1 to 4034.2]
  SARS-CoV-2 DB His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 DB His-50-N at Month 2-Total | 295.6 [1 to 1049.1] | 228.5 [1 to 1017.8] | 277.8 [1 to 1037.8] | 133.2 [1 to 1037.8] | 171.2 [1 to 1027.8] | 35.2 [1 to 720.2] | 205.8 [1 to 996] | 205.8 [1 to 946.2] | 211.2 [1 to 1022.8] | 133.2 [1 to 946.2] | 130.5 [1 to 913.1]
  SARS-CoV-2 DB His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 182 | 39 | 45 | 43 | 87 | 74
  SARS-CoV-2 DB His-50-Y at Month 0-Total | 846 [111.2 to 1581.2] | 1623.5 [587.8 to 3900.8] | 846 [185.2 to 1512.8] | 1392.2 [259.9 to 3686.8] | 1563.8 [468.1 to 3827.6] | 1936.8 [619.1 to 3975.9] | 1617 [398.4 to 4047.9] | 2579.5 [1091 to 4715.5] | 1696.2 [926.6 to 3524.1] | 1738.5 [356 to 4191] | 1982.8 [925.1 to 3346.4]
  SARS-CoV-2 DB His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 DB His-50-Y at Month 2-Total | 43.9 [1 to 482.1] | 346.5 [1 to 1136.4] | 205.8 [5.1 to 557.2] | 346.5 [1 to 857.4] | 277.8 [1 to 985.2] | 514.2 [33.5 to 1537.8] | 419.8 [1 to 2137.2] | 985.2 [194 to 1362.2] | 576.1 [154.6 to 1051.4] | 427.8 [21.5 to 1362.2] | 898.1 [421.6 to 1208.2]
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total: number analyzed (Participants) | 344 | 249 | 348 | 271 | 206 | 187 | 330 | 324 | 326 | 283 | 295
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total | 7626.2 [3266.3 to 14672.5] | 7312.8 [3108.5 to 14197.5] | 7626.2 [3330.2 to 14595.2] | 7569.5 [3347 to 14658.2] | 7366.4 [3346.1 to 14458.9] | 7442 [3104.1 to 14613.2] | 7378.5 [3137.7 to 14801.3] | 7378.5 [3035.7 to 14164.5] | 7790.1 [3101.9 to 14631.2] | 7442 [3315.1 to 14132] | 7941.5 [3072 to 14668.8]
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total | 1840 [474.7 to 4095.7] | 1827 [521 to 4059.2] | 1827 [415.8 to 4059.2] | 1404.5 [274.8 to 3572.8] | 1506 [273.8 to 3828.8] | 1482.5 [327.9 to 4294] | 1827 [463.9 to 4212.8] | 1506 [287.6 to 4049.4] | 2007.9 [403.6 to 4208.9] | 1404.5 [287.6 to 3397.5] | 1840 [379.4 to 4330.8]
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 182 | 39 | 45 | 43 | 86 | 74
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total | 5257.5 [519.5 to 9089.2] | 7812.2 [3193.9 to 14319.1] | 3931.8 [376.5 to 9487.2] | 7043.4 [2226.6 to 13076.2] | 7683 [3027.1 to 14193.2] | 7369.9 [3238.2 to 13901.4] | 7799 [3179.4 to 11897.2] | 8540.8 [4301.8 to 18738.2] | 4657.2 [3342.2 to 10291] | 7179.2 [1347.8 to 14683] | 5919 [3413.9 to 11878.8]
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total | 778.1 [1 to 1594.1] | 1404.5 [280.8 to 3625] | 1047.2 [408.9 to 2175.9] | 2177 [1060.2 to 4345.5] | 1787.8 [726.5 to 3893.8] | 1827 [485.5 to 3598.2] | 924.5 [1 to 3572.8] | 2177 [1385.5 to 3132.5] | 1184.4 [331.9 to 1486.1] | 2183 [1321.5 to 4205] | 1358.1 [593.5 to 2177.9]
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total: number analyzed (Participants) | 342 | 247 | 346 | 269 | 204 | 187 | 328 | 324 | 324 | 282 | 293
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total | 1770.9 [548.4 to 4375.2] | 1617.5 [524.4 to 4186.6] | 1739.8 [553.6 to 4362.8] | 1781 [701 to 4524.8] | 1670.5 [709.2 to 4355] | 1617.5 [534.6 to 4380.4] | 1670.5 [544.4 to 4286.1] | 1542.6 [513.1 to 4212.4] | 1703.5 [519.9 to 4369.1] | 1590.4 [538.3 to 4327.4] | 1660.2 [501.5 to 4376]
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total | 441.5 [5.5 to 1058.4] | 441.2 [1 to 1002] | 422 [1 to 1081.2] | 441.2 [1 to 1217.2] | 441.2 [1 to 1066] | 241.2 [1 to 1032.9] | 340.5 [1 to 1043.9] | 303 [1 to 1066] | 382.5 [1 to 1083.1] | 303 [1 to 1066] | 321.8 [1 to 1079.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 180 | 39 | 43 | 43 | 85 | 74
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total | 923 [20.5 to 1634.5] | 1957.2 [579 to 4535.8] | 650.2 [114.5 to 2615] | 1366.1 [166.3 to 3626.4] | 1634.5 [410.4 to 4225.4] | 1801.8 [513.1 to 4168.9] | 1184 [286.9 to 4187.2] | 2906.5 [1431.9 to 5722.5] | 1478.5 [706.6 to 2867.2] | 1917.8 [180 to 4153.8] | 1610.8 [730.2 to 2924]
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total | 75 [1 to 2548.4] | 267.2 [1 to 1624.6] | 143.2 [102.6 to 765.6] | 246.5 [48.9 to 942.5] | 267.2 [1 to 1037] | 595 [108.5 to 1088.8] | 610.2 [1 to 2049.8] | 771.8 [595 to 1002] | 405.8 [81.6 to 807.1] | 595 [7 to 1002] | 666.2 [173.4 to 1015.8]
  SARS-CoV-2 S1 C His-50-N at Month 0-Total: number analyzed (Participants) | 346 | 250 | 350 | 273 | 207 | 188 | 332 | 325 | 328 | 284 | 297
  SARS-CoV-2 S1 C His-50-N at Month 0-Total | 1957.5 [629.2 to 4714.1] | 1828.2 [513.6 to 4705.1] | 1870.2 [620.9 to 4651.9] | 1960.5 [784.8 to 4710.5] | 1954.5 [759.1 to 4726.4] | 1859.2 [582.8 to 4329.2] | 1859.2 [592.7 to 4706.1] | 1737.2 [511.5 to 4163.8] | 1859.2 [544.4 to 4694.1] | 1788 [613.9 to 4329.2] | 1833.5 [467 to 4715.2]
  SARS-CoV-2 S1 C His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1 C His-50-N at Month 2-Total | 657.5 [52.4 to 1488.5] | 662 [68.2 to 1331.2] | 616 [28.8 to 1479.5] | 414.2 [41.8 to 1535.5] | 489.8 [48.9 to 1525.5] | 235.8 [1 to 1174.1] | 489.8 [28.4 to 1322.2] | 352.5 [27.8 to 1264.5] | 552.9 [38.5 to 1368.3] | 352.5 [27.8 to 1322.2] | 442.6 [28.2 to 1288.9]
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 183 | 39 | 46 | 43 | 87 | 74
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total | 769.8 [43 to 1224.2] | 1804 [620 to 3977.2] | 764 [100.8 to 2152.5] | 1163.9 [249.6 to 3520] | 1649.9 [283.6 to 3782.9] | 1754.2 [456.4 to 4710.2] | 1365.8 [231 to 3437.1] | 2437.8 [1085.1 to 5691.8] | 1446 [621.9 to 3643.2] | 1960.5 [209.2 to 4737.8] | 1797.5 [741.1 to 3816.3]
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total | 164.5 [1 to 425.1] | 274.2 [8.5 to 1540.2] | 227.2 [183 to 862.5] | 781.2 [94.8 to 1157.5] | 616 [28.8 to 1196.2] | 957 [93.2 to 1835.2] | 1034.2 [68.2 to 2020.2] | 1200.5 [616 to 1658.2] | 681.2 [170.7 to 1287.1] | 690.5 [78 to 1547] | 1117.5 [243.1 to 1544.1]
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 343 | 247 | 348 | 271 | 205 | 186 | 329 | 322 | 326 | 281 | 295
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total | 8735.5 [3844.9 to 19163.8] | 8549.5 [3712.5 to 18041.2] | 8681.9 [3850.4 to 19160] | 8765.8 [4036.2 to 19141.5] | 8713.8 [4025.8 to 18259.8] | 8805.4 [3857.8 to 18034.1] | 8650 [3810 to 18958.5] | 7990.9 [3471.6 to 17828.5] | 9101.8 [3862.4 to 19167.5] | 8273.5 [3881.8 to 17676.2] | 9262.8 [3662.2 to 20130]
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total | 4900 [1970.3 to 10938.6] | 5013.2 [2166.2 to 10498.8] | 4119.8 [1952.5 to 10498.8] | 4254.2 [1952.5 to 8678] | 4964.2 [2019.1 to 11795.6] | 3503.5 [1849.2 to 10045.4] | 4368.2 [2004.8 to 10045.4] | 4254.2 [1918.2 to 10045.4] | 4311.2 [1948.8 to 10938.6] | 4119.8 [1925.6 to 10045.4] | 4187 [1941.4 to 10646.7]
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 20 | 97 | 163 | 182 | 39 | 46 | 42 | 87 | 73
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total | 6368 [2888.2 to 12087.5] | 8827 [3931.2 to 21444.8] | 7395.6 [2701.9 to 10007.4] | 6568.5 [2955 to 18021] | 8258.2 [3384.4 to 19087.8] | 8430.2 [3821.5 to 19205.6] | 8172 [3921.9 to 17855.4] | 15769.5 [5942.3 to 22000] | 5506.5 [3730.7 to 10496.1] | 8827 [2814 to 22000] | 6517.8 [3862.2 to 11943.5]
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total | 2803.2 [1525.2 to 4454.8] | 3715.2 [1454.1 to 8568.9] | 8445.8 [5613.2 to 9084] | 5013.2 [2391.2 to 10453.5] | 4119.8 [1898.8 to 9642.2] | 5260.2 [2074 to 10696] | 6527 [743.8 to 10696] | 4964.2 [3969.2 to 11944] | 5613.2 [3304.9 to 7430.6] | 5013.2 [2736.5 to 11944] | 6101.5 [3241.4 to 8133.9]
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total: number analyzed (Participants) | 346 | 250 | 350 | 273 | 207 | 188 | 332 | 325 | 328 | 284 | 297
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total | 4718.9 [2289.4 to 8954.2] | 4662.5 [2207.5 to 8345.1] | 4645 [2278.4 to 8763.1] | 4753 [2345.2 to 8839.8] | 4781.2 [2296.4 to 8438.8] | 4504.2 [2184.6 to 8824.9] | 4609 [2281.1 to 8537.1] | 4350 [2116 to 8313.2] | 4645 [2203.8 to 8824.9] | 4549.4 [2273 to 8537.1] | 4650.5 [2116 to 8918.8]
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total | 2095.1 [685.5 to 3415.7] | 2071.8 [547.8 to 2944.8] | 2048 [548 to 3405.5] | 1910 [456.5 to 2971.2] | 2048 [468.9 to 2958] | 1731 [510.1 to 2826.8] | 2048 [641.1 to 3138.1] | 1891 [543.4 to 2958] | 1979 [601.6 to 3415.7] | 1781.5 [543.4 to 2958] | 1836.2 [541.2 to 3380.4]
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 121 | 21 | 98 | 164 | 183 | 39 | 46 | 43 | 87 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total | 3164 [1113.8 to 4364.8] | 4366.2 [2277 to 9720.5] | 2512.2 [321.8 to 5041] | 3896 [1654.4 to 6961.9] | 4330.5 [2186 to 8894.9] | 4522.2 [2245 to 8542.2] | 3506 [1710.4 to 10522.6] | 6569.9 [3530.6 to 11213.2] | 3914.5 [2287.9 to 7157.9] | 4473 [1636.4 to 8731.8] | 3945 [2460.2 to 6991.4]
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total | 719.1 [1 to 1535.8] | 1748.2 [719.1 to 4054] | 2177 [1542.5 to 2305] | 2177 [1329.5 to 3375.6] | 2071.8 [946 to 3446.2] | 2211 [775.5 to 4123.8] | 2385.5 [202.8 to 3879] | 2739 [2254.8 to 4154.8] | 2192.4 [855.5 to 2288.8] | 2254.8 [947.5 to 4154.8] | 2209.4 [1238.6 to 2457]
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total: number analyzed (Participants) | 345 | 250 | 349 | 272 | 207 | 188 | 331 | 325 | 327 | 284 | 296
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total | 2900.2 [554 to 8391] | 2824.9 [454.8 to 8155.4] | 2865.8 [540.8 to 8208] | 3243.5 [732.4 to 8411.1] | 3017.8 [628.2 to 8396.5] | 2733.1 [516 to 8411.1] | 2890 [531.5 to 8396.5] | 2222.8 [411 to 7521.5] | 2839.2 [471.8 to 8266.8] | 2733.1 [521.2 to 8050.3] | 2698.6 [429.2 to 8393.8]
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total | 668.4 [128.8 to 1719.1] | 650.2 [119.8 to 1568.2] | 603.2 [126.8 to 1599.8] | 603 [119.8 to 1672.2] | 634 [128.1 to 1741.6] | 581 [83.8 to 1216.6] | 603.2 [113.2 to 1584] | 521.2 [36 to 1495] | 603.1 [119.4 to 1576.1] | 581 [113.2 to 1431.8] | 592.4 [118.8 to 1498.9]
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 120 | 21 | 98 | 163 | 182 | 39 | 45 | 43 | 86 | 74
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total | 394.8 [1.8 to 2021.8] | 2698.6 [516 to 7375.9] | 259.8 [6 to 4336.8] | 1502.9 [100.9 to 6241.9] | 2556 [263.5 to 6594] | 2839.1 [431.4 to 7203.9] | 1047 [140.9 to 4342.2] | 4505 [2362.8 to 10177.8] | 2308.5 [469.9 to 6322.8] | 2852.4 [9.8 to 6997] | 2941.8 [596.4 to 6333.1]
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total | 1 [1 to 467.8] | 349 [56.2 to 1743.8] | 59.5 [1 to 1413.2] | 809.2 [89 to 1527.8] | 581 [59.5 to 1502.8] | 686.5 [149 to 1811] | 581.8 [119.8 to 1672.2] | 1672.2 [903 to 1811] | 644.4 [3.2 to 1765.4] | 844 [199 to 1811] | 873.8 [46.8 to 2033]

50. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (IgA) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
Participants
  2019-nCoV S/293F-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  2019-nCoV S/293F-50-N at Month 0-Peru | 160 | 119 | 167 | 158 | 118 | 109 | 159 | 149 | 153 | 146 | 145
  2019-nCoV S/293F-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  2019-nCoV S/293F-50-N at Month 0-Total | 310 | 224 | 316 | 248 | 190 | 174 | 295 | 286 | 292 | 260 | 266
  2019-nCoV S/293F-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  2019-nCoV S/293F-50-N at Month 0-USA | 150 | 105 | 149 | 90 | 72 | 65 | 136 | 137 | 139 | 114 | 121
  2019-nCoV S/293F-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  2019-nCoV S/293F-50-N at Month 2-Peru | 25 | 20 | 28 | 26 | 19 | 20 | 28 | 24 | 26 | 25 | 25
  2019-nCoV S/293F-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  2019-nCoV S/293F-50-N at Month 2-Total | 80 | 63 | 81 | 56 | 44 | 46 | 74 | 77 | 79 | 65 | 73
  2019-nCoV S/293F-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  2019-nCoV S/293F-50-N at Month 2-USA | 55 | 43 | 53 | 30 | 25 | 26 | 46 | 53 | 53 | 40 | 48
  2019-nCoV S/293F-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  2019-nCoV S/293F-50-Y at Month 0-Peru | 7 | 48 | 0 | 9 | 49 | 58 | 8 | 18 | 14 | 21 | 22
  2019-nCoV S/293F-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  2019-nCoV S/293F-50-Y at Month 0-Total | 19 | 105 | 13 | 81 | 139 | 155 | 34 | 43 | 37 | 69 | 63
  2019-nCoV S/293F-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  2019-nCoV S/293F-50-Y at Month 0-USA | 12 | 57 | 13 | 72 | 90 | 97 | 26 | 25 | 23 | 48 | 41
  2019-nCoV S/293F-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  2019-nCoV S/293F-50-Y at Month 2-Peru | 3 | 8 | 0 | 2 | 9 | 8 | 0 | 4 | 2 | 3 | 3
  2019-nCoV S/293F-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  2019-nCoV S/293F-50-Y at Month 2-Total | 6 | 23 | 5 | 30 | 42 | 40 | 12 | 9 | 7 | 21 | 13
  2019-nCoV S/293F-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  2019-nCoV S/293F-50-Y at Month 2-USA | 3 | 15 | 5 | 28 | 33 | 32 | 12 | 5 | 5 | 18 | 10
  SARS-CoV-2 DB His-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 DB His-50-N at Month 0-Peru | 152 | 113 | 157 | 149 | 112 | 102 | 150 | 139 | 144 | 137 | 136
  SARS-CoV-2 DB His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 DB His-50-N at Month 0-Total | 267 | 191 | 274 | 220 | 168 | 146 | 255 | 242 | 250 | 222 | 226
  SARS-CoV-2 DB His-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 DB His-50-N at Month 0-USA | 115 | 78 | 117 | 71 | 56 | 44 | 105 | 103 | 106 | 85 | 90
  SARS-CoV-2 DB His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 DB His-50-N at Month 2-Peru | 21 | 17 | 23 | 22 | 16 | 17 | 23 | 19 | 22 | 20 | 22
  SARS-CoV-2 DB His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 DB His-50-N at Month 2-Total | 61 | 47 | 62 | 46 | 35 | 34 | 56 | 58 | 61 | 48 | 57
  SARS-CoV-2 DB His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 DB His-50-N at Month 2-USA | 40 | 30 | 39 | 24 | 19 | 17 | 33 | 39 | 39 | 28 | 35
  SARS-CoV-2 DB His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 DB His-50-Y at Month 0-Peru | 5 | 44 | 0 | 8 | 45 | 55 | 7 | 18 | 13 | 20 | 21
  SARS-CoV-2 DB His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 DB His-50-Y at Month 0-Total | 16 | 92 | 9 | 63 | 115 | 137 | 28 | 41 | 33 | 61 | 57
  SARS-CoV-2 DB His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 DB His-50-Y at Month 0-USA | 11 | 48 | 9 | 55 | 70 | 82 | 21 | 23 | 20 | 41 | 36
  SARS-CoV-2 DB His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 DB His-50-Y at Month 2-Peru | 2 | 6 | 0 | 1 | 7 | 6 | 0 | 4 | 1 | 3 | 1
  SARS-CoV-2 DB His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 DB His-50-Y at Month 2-Total | 4 | 18 | 3 | 19 | 30 | 31 | 9 | 7 | 4 | 17 | 8
  SARS-CoV-2 DB His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 DB His-50-Y at Month 2-USA | 2 | 12 | 3 | 18 | 23 | 25 | 9 | 3 | 3 | 14 | 7
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Peru | 159 | 118 | 164 | 155 | 117 | 107 | 155 | 147 | 153 | 142 | 145
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total | 301 | 215 | 305 | 238 | 181 | 165 | 285 | 282 | 285 | 249 | 258
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-USA | 142 | 97 | 141 | 83 | 64 | 58 | 130 | 135 | 132 | 107 | 113
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Peru | 27 | 22 | 30 | 29 | 21 | 21 | 29 | 26 | 29 | 26 | 28
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total | 73 | 57 | 74 | 54 | 42 | 40 | 67 | 71 | 73 | 59 | 67
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-USA | 46 | 35 | 44 | 25 | 21 | 19 | 38 | 45 | 44 | 33 | 39
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Peru | 5 | 46 | 0 | 9 | 47 | 57 | 9 | 17 | 11 | 22 | 19
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total | 21 | 107 | 17 | 84 | 141 | 157 | 37 | 40 | 37 | 73 | 64
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-USA | 16 | 61 | 17 | 75 | 94 | 100 | 28 | 23 | 26 | 51 | 45
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Peru | 3 | 8 | 0 | 1 | 9 | 9 | 1 | 4 | 1 | 4 | 2
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total | 6 | 22 | 5 | 25 | 37 | 39 | 12 | 8 | 6 | 20 | 12
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-USA | 3 | 14 | 5 | 24 | 28 | 30 | 11 | 4 | 5 | 16 | 10
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Peru | 162 | 119 | 169 | 160 | 118 | 110 | 161 | 151 | 154 | 148 | 146
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total | 314 | 226 | 319 | 251 | 191 | 176 | 299 | 290 | 294 | 264 | 268
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-USA | 152 | 107 | 150 | 91 | 73 | 66 | 138 | 139 | 140 | 116 | 122
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Peru | 26 | 21 | 30 | 28 | 20 | 22 | 30 | 26 | 28 | 27 | 27
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total | 82 | 65 | 83 | 58 | 45 | 49 | 77 | 79 | 82 | 67 | 76
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-USA | 56 | 44 | 53 | 30 | 25 | 27 | 47 | 53 | 54 | 40 | 49
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Peru | 7 | 50 | 0 | 9 | 51 | 59 | 8 | 18 | 15 | 21 | 23
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total | 19 | 107 | 14 | 82 | 142 | 157 | 34 | 43 | 39 | 69 | 65
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-USA | 12 | 57 | 14 | 73 | 91 | 98 | 26 | 25 | 24 | 48 | 42
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Peru | 4 | 9 | 0 | 2 | 10 | 8 | 0 | 4 | 2 | 3 | 3
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total | 6 | 23 | 5 | 30 | 43 | 39 | 11 | 9 | 6 | 21 | 12
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-USA | 2 | 14 | 5 | 28 | 33 | 31 | 11 | 5 | 4 | 18 | 9
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 S1 C His-50-N at Month 0-Peru | 160 | 119 | 166 | 158 | 118 | 109 | 158 | 148 | 152 | 146 | 144
  SARS-CoV-2 S1 C His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S1 C His-50-N at Month 0-Total | 304 | 219 | 309 | 244 | 186 | 169 | 288 | 280 | 284 | 256 | 258
  SARS-CoV-2 S1 C His-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 S1 C His-50-N at Month 0-USA | 144 | 100 | 143 | 86 | 68 | 60 | 130 | 132 | 132 | 110 | 114
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S1 C His-50-N at Month 2-Peru | 25 | 20 | 27 | 25 | 19 | 20 | 27 | 23 | 25 | 24 | 25
  SARS-CoV-2 S1 C His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1 C His-50-N at Month 2-Total | 77 | 61 | 77 | 54 | 43 | 43 | 70 | 72 | 75 | 60 | 70
  SARS-CoV-2 S1 C His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S1 C His-50-N at Month 2-USA | 52 | 41 | 50 | 29 | 24 | 23 | 43 | 49 | 50 | 36 | 45
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 S1 C His-50-Y at Month 0-Peru | 6 | 47 | 0 | 8 | 48 | 57 | 8 | 18 | 14 | 20 | 22
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total | 18 | 103 | 13 | 78 | 136 | 153 | 34 | 42 | 38 | 66 | 64
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 S1 C His-50-Y at Month 0-USA | 12 | 56 | 13 | 70 | 88 | 96 | 26 | 24 | 24 | 46 | 42
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S1 C His-50-Y at Month 2-Peru | 2 | 7 | 0 | 2 | 8 | 7 | 0 | 4 | 2 | 3 | 2
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total | 4 | 20 | 4 | 27 | 38 | 38 | 11 | 9 | 6 | 21 | 11
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S1 C His-50-Y at Month 2-USA | 2 | 13 | 4 | 25 | 30 | 31 | 11 | 5 | 4 | 18 | 9
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Peru | 104 | 78 | 107 | 104 | 77 | 67 | 101 | 90 | 102 | 90 | 97
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total | 163 | 114 | 165 | 140 | 105 | 85 | 151 | 135 | 156 | 124 | 140
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-USA | 59 | 36 | 58 | 36 | 28 | 18 | 50 | 45 | 54 | 34 | 43
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Peru | 9 | 7 | 11 | 11 | 7 | 6 | 11 | 7 | 10 | 9 | 10
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total | 29 | 21 | 29 | 22 | 16 | 12 | 25 | 25 | 28 | 20 | 26
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-USA | 20 | 14 | 18 | 11 | 9 | 6 | 14 | 18 | 18 | 11 | 16
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Peru | 3 | 29 | 0 | 3 | 30 | 40 | 6 | 17 | 5 | 17 | 10
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total | 5 | 54 | 3 | 28 | 63 | 83 | 17 | 33 | 12 | 44 | 28
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-USA | 2 | 25 | 3 | 25 | 33 | 43 | 11 | 16 | 7 | 27 | 18
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Peru | 2 | 4 | 0 | 0 | 4 | 5 | 0 | 4 | 1 | 2 | 1
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total | 2 | 10 | 2 | 9 | 15 | 19 | 6 | 6 | 3 | 11 | 5
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-USA | 0 | 6 | 2 | 9 | 11 | 14 | 6 | 2 | 2 | 9 | 4
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru: number analyzed (Participants) | 171 | 126 | 178 | 169 | 125 | 114 | 169 | 160 | 163 | 153 | 155
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Peru | 157 | 116 | 163 | 154 | 115 | 106 | 155 | 145 | 150 | 142 | 142
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total | 297 | 214 | 303 | 239 | 182 | 165 | 282 | 272 | 280 | 247 | 254
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA: number analyzed (Participants) | 177 | 125 | 174 | 105 | 83 | 75 | 165 | 166 | 167 | 132 | 144
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-USA | 140 | 98 | 140 | 85 | 67 | 59 | 127 | 127 | 130 | 105 | 112
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Peru | 22 | 19 | 24 | 23 | 18 | 18 | 24 | 20 | 23 | 21 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total | 75 | 60 | 75 | 52 | 42 | 43 | 68 | 70 | 74 | 59 | 69
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-USA | 53 | 41 | 51 | 29 | 24 | 25 | 44 | 50 | 51 | 38 | 46
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 64 | 9 | 18 | 15 | 25 | 23
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Peru | 6 | 47 | 0 | 9 | 48 | 57 | 8 | 18 | 13 | 21 | 21
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total | 18 | 101 | 12 | 76 | 133 | 150 | 33 | 43 | 35 | 68 | 61
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA: number analyzed (Participants) | 18 | 70 | 21 | 90 | 112 | 120 | 30 | 29 | 28 | 63 | 51
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-USA | 12 | 54 | 12 | 67 | 85 | 93 | 25 | 25 | 22 | 47 | 40
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Peru | 2 | 5 | 0 | 1 | 6 | 6 | 0 | 4 | 1 | 3 | 1
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total | 4 | 19 | 4 | 27 | 37 | 36 | 11 | 9 | 5 | 20 | 10
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-USA | 2 | 14 | 4 | 26 | 31 | 30 | 11 | 5 | 4 | 17 | 9
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru: number analyzed (Participants) | 135 | 95 | 140 | 134 | 94 | 84 | 133 | 125 | 125 | 119 | 119
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Peru | 120 | 85 | 124 | 118 | 84 | 74 | 118 | 109 | 110 | 107 | 104
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total: number analyzed (Participants) | 254 | 174 | 259 | 206 | 149 | 130 | 248 | 236 | 233 | 204 | 214
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total | 195 | 128 | 198 | 158 | 112 | 96 | 191 | 174 | 173 | 157 | 158
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA: number analyzed (Participants) | 119 | 79 | 119 | 72 | 55 | 46 | 115 | 111 | 108 | 85 | 95
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-USA | 75 | 43 | 74 | 40 | 28 | 22 | 73 | 65 | 63 | 50 | 54
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru: number analyzed (Participants) | 30 | 24 | 34 | 32 | 23 | 24 | 33 | 30 | 32 | 30 | 31
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Peru | 21 | 18 | 23 | 22 | 17 | 17 | 23 | 19 | 22 | 20 | 22
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total | 57 | 45 | 58 | 43 | 34 | 31 | 52 | 52 | 55 | 44 | 51
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA: number analyzed (Participants) | 62 | 49 | 59 | 33 | 28 | 31 | 54 | 61 | 60 | 45 | 55
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-USA | 36 | 27 | 35 | 21 | 17 | 14 | 29 | 33 | 33 | 24 | 29
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru: number analyzed (Participants) | 5 | 45 | 0 | 6 | 46 | 56 | 7 | 15 | 15 | 21 | 21
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Peru | 4 | 39 | 0 | 6 | 40 | 50 | 6 | 15 | 14 | 17 | 20
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total: number analyzed (Participants) | 21 | 101 | 16 | 69 | 126 | 145 | 27 | 39 | 42 | 71 | 61
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total | 12 | 79 | 9 | 49 | 95 | 111 | 16 | 33 | 34 | 50 | 49
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA: number analyzed (Participants) | 16 | 56 | 16 | 63 | 80 | 89 | 20 | 24 | 27 | 50 | 40
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-USA | 8 | 40 | 9 | 43 | 55 | 61 | 10 | 18 | 20 | 33 | 29
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru: number analyzed (Participants) | 4 | 10 | 0 | 2 | 11 | 10 | 1 | 4 | 2 | 4 | 3
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Peru | 2 | 5 | 0 | 1 | 6 | 6 | 0 | 4 | 1 | 3 | 1
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total | 3 | 15 | 2 | 17 | 26 | 29 | 8 | 8 | 5 | 16 | 9
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA: number analyzed (Participants) | 4 | 17 | 7 | 33 | 38 | 35 | 12 | 5 | 6 | 21 | 11
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-USA | 1 | 10 | 2 | 16 | 20 | 23 | 8 | 4 | 4 | 13 | 8

51. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgA) by Region and Comorbidity Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgA) at Visit 1, 2, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
MFI
  2019-nCoV S/293F-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  2019-nCoV S/293F-50-N at Month 0-Total | 7557.6 [2929.8 to 14389.8] | 6875.2 [2794.2 to 14286.1] | 7658 [3024.7 to 14622.6] | 8354.6 [3296.6 to 16184.8] | 8285 [3423.6 to 16183.2] | 7325.5 [2802.2 to 15131.5] | 7542.5 [2767.1 to 14875.8] | 6569.8 [2615.1 to 13142.6] | 7557.6 [2768.4 to 14875.8] | 6934.2 [2802.2 to 13813] | 7548.5 [2750.8 to 15093.5]
  2019-nCoV S/293F-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  2019-nCoV S/293F-50-N at Month 2-Total | 3795.1 [1839.1 to 7132.3] | 3154.8 [1724.5 to 6588] | 3758 [1724.5 to 7246.2] | 3951.5 [1877.2 to 7265.5] | 3758 [1882.1 to 7158.8] | 3301.5 [1805.8 to 6779.5] | 3758 [1645.5 to 7147.6] | 3227.5 [1546.9 to 7048.4] | 3618 [1685 to 7132.3] | 3136.2 [1625.9 to 6746.5] | 3839.1 [1765.1 to 7162.9]
  2019-nCoV S/293F-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  2019-nCoV S/293F-50-Y at Month 0-Total | 2914.2 [796.8 to 8142] | 7904.1 [2678.6 to 13718] | 1643.2 [190.2 to 4629.8] | 5132.5 [1634.2 to 8695.9] | 5966 [1700.5 to 11838.5] | 7152 [2636.4 to 12849.1] | 5832.2 [2604.6 to 8963] | 9327.8 [5674.1 to 19226.1] | 4969 [2559.5 to 8537.9] | 7639.2 [1589.6 to 14543.4] | 6037.8 [2787.1 to 10148.3]
  2019-nCoV S/293F-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  2019-nCoV S/293F-50-Y at Month 2-Total | 1780.2 [718.4 to 4146.1] | 5632.8 [1242.1 to 9509.2] | 1923.2 [643.4 to 3306.8] | 3154.8 [1499.8 to 5749.1] | 3227.5 [1472.2 to 7117] | 3832.2 [1527.2 to 7392.8] | 2658.2 [1527.2 to 7044.8] | 6300 [3112.8 to 10458.8] | 2329.2 [800.1 to 5488.9] | 6300 [1566.5 to 9431.2] | 2749.2 [1218.1 to 6122.8]
  229E-RBD-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  229E-RBD-50-N at Month 0-Total | 524.4 [301.6 to 980] | 521.2 [291.9 to 903.4] | 533.2 [317.9 to 970.4] | 546.2 [334.3 to 966.9] | 556.2 [331.8 to 914.2] | 487.5 [325.2 to 898] | 517.5 [304.8 to 943.1] | 506.6 [291.7 to 916.1] | 513 [299.2 to 933.8] | 520.5 [298 to 925] | 504 [317.1 to 930.9]
  229E-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  229E-RBD-50-N at Month 2-Total | 339.6 [217.4 to 715.7] | 321 [202.8 to 649.5] | 341 [219 to 708.8] | 321 [205.2 to 708.8] | 321 [203.5 to 784.2] | 299.2 [204.8 to 494.5] | 338.2 [219.1 to 670.2] | 341 [214.1 to 722.6] | 339.6 [211.7 to 715.7] | 313.5 [207.2 to 663.2] | 329.9 [210.1 to 697.8]
  229E-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  229E-RBD-50-Y at Month 0-Total | 419.5 [259.8 to 808.5] | 510.4 [318.6 to 1026.1] | 320.8 [222.2 to 673.8] | 466.8 [241.9 to 879] | 487 [276.5 to 979] | 582.4 [288.4 to 1055.2] | 525.5 [293.6 to 1076.1] | 725.2 [345.5 to 1233.2] | 624.8 [300.1 to 1056.8] | 520 [300.8 to 1059.4] | 582.4 [288.5 to 1040.5]
  229E-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  229E-RBD-50-Y at Month 2-Total | 402.4 [260.5 to 561.1] | 382.8 [303.9 to 807.5] | 445 [209.8 to 699.8] | 445 [240.2 to 713.8] | 382.2 [242 to 691] | 480.5 [295.8 to 938] | 445 [195.8 to 909.8] | 480.5 [295.8 to 700] | 394.6 [283.2 to 692.4] | 459.2 [295.8 to 1034.8] | 490.1 [307.9 to 1342.4]
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  HCoV-229E S1S2 ECD His-50-N at Month 0-Total | 463.1 [229.6 to 989.9] | 429.5 [218.2 to 876] | 469.1 [239.5 to 999.6] | 467.2 [249.6 to 1023.6] | 439.5 [232.7 to 916.6] | 451.8 [220 to 888.2] | 463.1 [221.3 to 954.7] | 467.2 [231.6 to 972.4] | 465.6 [226.7 to 954.7] | 453.8 [220 to 986.5] | 465.8 [235.1 to 935.4]
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-229E S1S2 ECD His-50-N at Month 2-Total | 465.8 [174.8 to 984.4] | 447 [176 to 885.5] | 533.2 [190.2 to 1058.2] | 486.5 [187.5 to 1095] | 483 [203.4 to 1133.1] | 402 [166.9 to 873.8] | 483 [188.9 to 915.8] | 482.8 [173.5 to 1037.4] | 484.8 [184.6 to 973.9] | 483 [166.9 to 967.5] | 482.9 [178.9 to 912.2]
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  HCoV-229E S1S2 ECD His-50-Y at Month 0-Total | 603.8 [286.8 to 954.5] | 588.1 [246.6 to 1187.1] | 286.8 [128.5 to 491.2] | 436.8 [159.1 to 889] | 492.8 [199.5 to 1059] | 472.5 [238.1 to 1052.9] | 567.5 [267.9 to 1090.8] | 465.5 [230.1 to 1041.9] | 508.8 [260 to 1061.6] | 480.1 [275 to 959.3] | 456.9 [183.8 to 1091.8]
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-229E S1S2 ECD His-50-Y at Month 2-Total | 822.8 [573.6 to 1036.1] | 698 [198 to 1529.5] | 303.2 [137.8 to 633.1] | 482.8 [227.1 to 915.8] | 603.8 [176 to 918.5] | 670.5 [282.2 to 1320.2] | 786 [149.8 to 1699.8] | 614.2 [293.5 to 843.5] | 608.1 [253.9 to 1556.9] | 561 [284.2 to 1250.2] | 791.8 [289 to 1697.1]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 0-Total | 1381 [613 to 3349.1] | 1351.8 [601.5 to 3152.2] | 1451.1 [628.4 to 3349.1] | 1417.8 [621.6 to 3305] | 1433.1 [613 to 3206.4] | 1240 [607 to 2576.8] | 1309.2 [608.9 to 2958.9] | 1309.2 [607.4 to 3080.4] | 1398.9 [608.9 to 3305] | 1351.8 [614 to 2959.8] | 1418.5 [617.4 to 3281]
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-HKU1 N5 S1S2 ECD His-50-N at Month 2-Total | 1281.4 [609.1 to 3178.1] | 1266.5 [528.5 to 3260] | 1462.2 [615.8 to 3150.8] | 1582 [459.5 to 3499.2] | 1582 [434.1 to 4022.1] | 1296.2 [561.1 to 2817] | 1226.5 [604 to 2817] | 1296.2 [561.1 to 3205.4] | 1478.1 [575.1 to 3178.1] | 1462.2 [602.4 to 3123.6] | 1379.2 [595.7 to 3132.2]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 0-Total | 1310 [646.8 to 2772.2] | 1416.4 [690.2 to 3500.2] | 809.2 [499 to 1310] | 1310 [605.2 to 3067.9] | 1350.2 [626 to 3168.5] | 1563.2 [651.9 to 3921.3] | 3089 [976.8 to 5111.9] | 1754 [695.6 to 4131.2] | 1348 [697.5 to 2720.9] | 1440.9 [621.6 to 4846.4] | 1297.5 [593.8 to 3024.2]
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-HKU1 N5 S1S2 ECD His-50-Y at Month 2-Total | 1340.1 [874.9 to 1979.1] | 1296.2 [779.9 to 2465] | 847.5 [551.6 to 1376.6] | 1009.5 [821.5 to 2090.6] | 1266.5 [798.2 to 2437.5] | 1266.5 [619 to 3471.5] | 2905.5 [615.8 to 4816.8] | 1266.5 [1010 to 1888.2] | 811.8 [653.6 to 1193.1] | 1255.2 [619 to 3150.8] | 963.6 [650.9 to 3450]
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  HCoV-NL63 S1S2 ECD His-50-N at Month 0-Total | 83.9 [30.4 to 186] | 84.5 [30.9 to 186] | 86.1 [30.9 to 195.9] | 80.5 [30 to 185.6] | 83.8 [29.9 to 186.1] | 76.5 [30.5 to 177.2] | 80.5 [30 to 189.8] | 86.1 [30.5 to 188] | 79.4 [30.1 to 184.4] | 83.2 [31.2 to 184.2] | 78.8 [30.5 to 181.4]
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 91 | 72 | 92 | 64 | 50 | 54 | 85 | 89 | 91 | 74 | 85
  HCoV-NL63 S1S2 ECD His-50-N at Month 2-Total | 90.8 [40.2 to 172] | 90.8 [41 to 194.6] | 91.4 [47.1 to 187.1] | 88.4 [49.1 to 190.3] | 93.2 [48.2 to 221.4] | 84.2 [38.2 to 164.8] | 86.8 [38.8 to 186.5] | 86.8 [41.8 to 167.8] | 90.8 [43.4 to 187.8] | 89.9 [45.5 to 183.9] | 89 [38.8 to 167.8]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  HCoV-NL63 S1S2 ECD His-50-Y at Month 0-Total | 94 [56 to 214.8] | 85.9 [31.3 to 203.8] | 69.8 [44.5 to 147.2] | 94.5 [46.1 to 213.6] | 86 [32.5 to 196.2] | 92.1 [32.2 to 209.6] | 128.2 [46.8 to 188.5] | 73 [38.4 to 209.9] | 105 [51.5 to 299.9] | 86.9 [30.8 to 205.7] | 95 [33 to 290.1]
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 7 | 26 | 6 | 34 | 48 | 44 | 13 | 9 | 7 | 24 | 13
  HCoV-NL63 S1S2 ECD His-50-Y at Month 2-Total | 65.2 [54.2 to 210.6] | 80.5 [52.9 to 152.1] | 33.6 [9.9 to 70.2] | 91.4 [37.1 to 164.8] | 80.4 [38.2 to 158.4] | 93.2 [51.9 to 190.3] | 98 [82 to 167.8] | 121.2 [89 to 195.5] | 79 [49.1 to 96.2] | 88.6 [36.2 to 159.5] | 94.5 [57 to 194.2]
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  HCoV-OC43 S1S2 ECD His-50-N at Month 0-Total | 3141.6 [1489.9 to 6449.9] | 2869.5 [1365.4 to 6218.6] | 3285.8 [1553.4 to 6457.3] | 3177.8 [1476.4 to 6430] | 2926.1 [1371.4 to 6366.1] | 2708.8 [1470.5 to 5545.2] | 3002.4 [1454 to 6082] | 3069.2 [1471.3 to 6185] | 3141.6 [1518.5 to 6368.2] | 3213.8 [1491.8 to 6056.5] | 3270.5 [1620.4 to 6307.6]
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HCoV-OC43 S1S2 ECD His-50-N at Month 2-Total | 2630.5 [1201.6 to 6157.4] | 2467 [1071.2 to 6169.2] | 2895.8 [1205.8 to 6153.5] | 2701 [1066.5 to 6424] | 2625.5 [870.6 to 6587.6] | 3008.5 [1197.5 to 5088.8] | 2625.5 [1197.5 to 5397.8] | 2701 [1197.5 to 6092.6] | 2952.1 [1201.6 to 6157.4] | 2895.8 [1207.1 to 5601] | 2952.1 [1206.4 to 5986.2]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  HCoV-OC43 S1S2 ECD His-50-Y at Month 0-Total | 3285.8 [1675.5 to 5733] | 3430.2 [1817.9 to 6647.2] | 2578.2 [972.2 to 3085.8] | 3085.8 [1603.4 to 6145.2] | 3274.5 [1675.5 to 6222.8] | 3515.8 [1548.5 to 6838.9] | 4889.5 [2332.2 to 9436.5] | 3706.2 [1825.6 to 7798.9] | 3356.8 [1364.1 to 6156.6] | 3097.1 [1587.2 to 7991.9] | 2747.6 [1138.3 to 6393]
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HCoV-OC43 S1S2 ECD His-50-Y at Month 2-Total | 3165.8 [2112.6 to 5410.4] | 3008.5 [2083.9 to 4999.2] | 2402.5 [1052.1 to 4075.6] | 2436 [1403.8 to 5873.5] | 2701 [1407 to 5308.8] | 2467 [1323 to 6968] | 5715.2 [2030 to 8553.8] | 1773.8 [1486.2 to 4229.5] | 2419.2 [1884.1 to 3397.9] | 2436 [1123 to 7176.2] | 2419.2 [1207 to 6396.4]
  HKU1-RBD-50-N at Month 0-Total: number analyzed (Participants) | 347 | 250 | 351 | 274 | 208 | 189 | 333 | 325 | 330 | 284 | 299
  HKU1-RBD-50-N at Month 0-Total | 458.5 [287 to 820.2] | 460.9 [286.6 to 817.4] | 473.5 [288.4 to 832.6] | 484.1 [292.9 to 848.5] | 491.5 [301.6 to 833.6] | 476.8 [281.5 to 805.2] | 448.8 [271 to 832.8] | 453 [271.2 to 809] | 449.6 [273.6 to 808.1] | 481.6 [299 to 816.7] | 453 [273.6 to 797.6]
  HKU1-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  HKU1-RBD-50-N at Month 2-Total | 403.9 [236 to 738.8] | 403.2 [210.8 to 774.5] | 403.2 [236 to 767.5] | 409.2 [239 to 847] | 442.8 [239.9 to 943.2] | 358.2 [173 to 758.1] | 376.2 [202.9 to 739.1] | 393 [217.1 to 758.1] | 395.2 [220.3 to 753.4] | 404.5 [229.8 to 777.9] | 388.4 [213.9 to 726]
  HKU1-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 98 | 164 | 183 | 39 | 47 | 42 | 88 | 73
  HKU1-RBD-50-Y at Month 0-Total | 475.5 [269 to 1433] | 457.8 [273.6 to 856.4] | 362.5 [223.2 to 833] | 405.2 [236.2 to 767.8] | 414.8 [260.8 to 832.8] | 447.2 [281.1 to 877.2] | 567.8 [328.9 to 826.6] | 514.2 [327.2 to 1603.5] | 547.9 [325.2 to 1146.7] | 387.2 [243.1 to 874.1] | 520 [306.2 to 1071.5]
  HKU1-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  HKU1-RBD-50-Y at Month 2-Total | 484.2 [168.4 to 758.4] | 404.5 [282.5 to 712.5] | 481 [209.2 to 673.9] | 403.2 [202.9 to 620.4] | 383.8 [210.8 to 622.5] | 442.8 [291.5 to 729.5] | 536.2 [421.8 to 787.5] | 536.2 [397.5 to 729.2] | 577.2 [439.8 to 744] | 403.2 [236 to 587.5] | 577.2 [389.1 to 1098.4]
  NL63-RBD-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  NL63-RBD-50-N at Month 0-Total | 1211.6 [675.3 to 2475.4] | 1191.2 [651 to 2317.8] | 1224.5 [699.7 to 2506.1] | 1211.6 [703.9 to 2231.5] | 1213.1 [689.3 to 2508.4] | 1191.2 [681.2 to 2022.5] | 1192.4 [640.8 to 2311.5] | 1197.6 [663.4 to 2556.6] | 1235 [723.1 to 2493.1] | 1217 [657.5 to 2302.5] | 1241 [747.5 to 2322.1]
  NL63-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  NL63-RBD-50-N at Month 2-Total | 1096.9 [607 to 2441.9] | 1048.8 [604 to 2371] | 1186.8 [637.8 to 2654.5] | 1269.5 [676 to 2654.5] | 1289.2 [663.4 to 3099.6] | 1128.2 [526.5 to 2825.1] | 1185.8 [632.1 to 2679.5] | 1225.2 [643 to 2825.1] | 1206 [669.1 to 2441.9] | 1186.8 [594 to 2310.1] | 1186.2 [679.2 to 2243.3]
  NL63-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  NL63-RBD-50-Y at Month 0-Total | 1619 [967.8 to 3627] | 1351.5 [784.4 to 2656.1] | 1170.5 [584.2 to 2664] | 1288.5 [628.6 to 3303.4] | 1241 [699.5 to 2510.8] | 1282.5 [712.1 to 2879.1] | 1708.2 [1000.1 to 4031.9] | 1582.5 [752.9 to 2322.1] | 917.5 [589.2 to 2738.8] | 1258 [745.6 to 3099.6] | 1075.1 [596.2 to 3270.6]
  NL63-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  NL63-RBD-50-Y at Month 2-Total | 1627.4 [1262 to 3635] | 1467.5 [737.9 to 3210.5] | 1126.5 [726.9 to 2826.1] | 942.5 [594 to 2578.9] | 1067.2 [626.5 to 1800] | 1186.8 [712.2 to 2371] | 1566.2 [1033.8 to 2249.2] | 1048.8 [626.5 to 1454.8] | 867.2 [547.8 to 4077.3] | 1185.8 [712.2 to 3291.2] | 1402.5 [590 to 4310.4]
  OC43-RBD-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  OC43-RBD-50-N at Month 0-Total | 485.8 [289.6 to 993.6] | 459.5 [270.9 to 884.5] | 497.8 [296.1 to 1034] | 489.9 [297.8 to 884.9] | 469.9 [288.9 to 884.1] | 477.2 [267 to 990.2] | 482.6 [276.2 to 1009.1] | 484.5 [280.1 to 987.1] | 479.1 [289.8 to 1020.9] | 500 [268 to 1037.8] | 484.2 [283.4 to 1005.2]
  OC43-RBD-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  OC43-RBD-50-N at Month 2-Total | 494.6 [272.7 to 1033.3] | 471 [252 to 987.2] | 492 [276.8 to 1042.5] | 492 [283.8 to 1030.2] | 492 [281.6 to 1036.9] | 423.5 [246.4 to 1132.4] | 471 [251 to 979] | 497.2 [257.4 to 1067.1] | 484.4 [260.1 to 1042.8] | 477.8 [269.8 to 1252.9] | 484.4 [248.8 to 1019.5]
  OC43-RBD-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  OC43-RBD-50-Y at Month 0-Total | 571.2 [303 to 1478.8] | 556.9 [329.9 to 1173.3] | 457.5 [215 to 977.8] | 524.2 [268.6 to 1151.4] | 527 [290 to 1114] | 510.1 [300.4 to 1067.4] | 598 [372.8 to 1044] | 673 [330.2 to 1216.8] | 576 [295.5 to 1034.8] | 469.6 [314.2 to 906.7] | 510.1 [313.1 to 1103.6]
  OC43-RBD-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  OC43-RBD-50-Y at Month 2-Total | 570.5 [308.1 to 1176.1] | 708.8 [313.6 to 1521.4] | 699.8 [168.9 to 811.6] | 552.2 [222.1 to 978.5] | 497.2 [247.8 to 914.5] | 699.8 [293.5 to 1016.8] | 920.8 [598.8 to 1271.2] | 491 [451.2 to 805] | 756.9 [593.8 to 940.1] | 708.8 [276 to 941.2] | 756.9 [350.2 to 1626.3]
  SARS-CoV-2 DB His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 DB His-50-N at Month 0-Total | 2970.9 [985.9 to 7455.9] | 2799.5 [935 to 7520] | 3017.9 [1062.2 to 7505.8] | 3695.4 [1232.6 to 8754.6] | 3567.9 [1267.2 to 8539.2] | 2997.5 [956.5 to 8169.8] | 3041.8 [934.6 to 7614.7] | 2583 [773.8 to 7069.1] | 2923.6 [908.6 to 7470.1] | 2882.5 [1011.2 to 7591.2] | 3038.2 [880.9 to 7700]
  SARS-CoV-2 DB His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 DB His-50-N at Month 2-Total | 1792.5 [547.2 to 3940.6] | 1634.5 [498 to 3583.2] | 1828.5 [596.8 to 3889] | 1916.8 [613.2 to 4095.5] | 1909.5 [547.4 to 3863.2] | 1360.8 [441.9 to 3133.9] | 1828.5 [483.5 to 3724.5] | 1561.5 [534.8 to 3597.4] | 1824.8 [587.5 to 3850.4] | 1433.2 [597 to 3133.9] | 1865.2 [522.2 to 3781]
  SARS-CoV-2 DB His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 DB His-50-Y at Month 0-Total | 1625.8 [569.5 to 2977] | 2914.4 [900.7 to 6144.4] | 583.2 [326.5 to 2002.5] | 1765.2 [500.9 to 3842.6] | 2041.2 [610.8 to 5292.5] | 2737.1 [790.4 to 6520.1] | 1532.8 [637.6 to 5278.5] | 4335.2 [2076.8 to 9723.9] | 1765.2 [977.6 to 5405.9] | 2495.6 [371.2 to 5380.9] | 2082.6 [1009.9 to 5510.9]
  SARS-CoV-2 DB His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 DB His-50-Y at Month 2-Total | 1048.4 [527.4 to 2301.8] | 2167.2 [632.4 to 5276.4] | 651.5 [438.9 to 1636] | 1159.2 [454.8 to 2832.1] | 1634.5 [559.8 to 3183] | 1828.5 [651.5 to 4926.5] | 1433.2 [709.8 to 4926.5] | 3183.2 [1949.8 to 7526] | 1143 [443.3 to 3432.1] | 2579.5 [448.5 to 5104.5] | 1361.2 [610.8 to 4612.3]
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 Nucleoprotein His-50-N at Month 0-Total | 2068.6 [606.9 to 5988.2] | 2155.8 [594.4 to 6034] | 1993.4 [596.1 to 5864.7] | 2203.2 [781.9 to 6285.1] | 2453.6 [798.8 to 6563.8] | 1929 [553.8 to 5346] | 1964.6 [521.1 to 5898.6] | 1771 [521.1 to 5312.6] | 2015.6 [600.8 to 5794.8] | 1929 [563 to 5746.2] | 1994 [558.4 to 5594.8]
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 Nucleoprotein His-50-N at Month 2-Total | 859.8 [421.5 to 1999.6] | 835.8 [425.8 to 2017.2] | 835.8 [425.8 to 1993.8] | 870.2 [431.2 to 2536.5] | 870.2 [429.1 to 2490.9] | 654.2 [285.5 to 1388.9] | 849.2 [386.6 to 1956.5] | 773.5 [405.2 to 1774.2] | 842.5 [426.7 to 2058.1] | 778.5 [417.2 to 1774.2] | 780.5 [426.1 to 1945.4]
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 0-Total | 520.8 [354.2 to 1115.2] | 1467.9 [490.6 to 4494.6] | 416.2 [323.2 to 2175.8] | 1115.2 [358.1 to 3474.4] | 1358 [416.2 to 3924.2] | 1905.1 [514.5 to 6368.9] | 1308.5 [849 to 4181.8] | 3375.5 [1170.4 to 9410.9] | 1126.8 [428.9 to 4308.6] | 1899.5 [356.7 to 6107.2] | 1553.8 [462 to 6273.2]
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 Nucleoprotein His-50-Y at Month 2-Total | 589.8 [456.8 to 1429.9] | 876.2 [421.4 to 1747.1] | 1491.8 [410.8 to 2433.4] | 773.5 [297.5 to 1529] | 782.5 [371.5 to 1566.2] | 1427.5 [447.8 to 3236] | 567.8 [520 to 2017.2] | 2332.5 [876.2 to 3236] | 978.6 [303 to 1598.6] | 1427.5 [431.2 to 2332.5] | 1406 [432.6 to 3156]
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 0-Total | 3082.4 [1055.1 to 7041.6] | 2691.8 [1040 to 6749] | 3168.6 [1084.2 to 7416.5] | 3524.9 [1171.8 to 8455.2] | 3351.5 [1164.6 to 8437.3] | 3151.2 [1049.8 to 8212.8] | 3168.6 [1002.5 to 7701.1] | 2649.5 [877.6 to 6580.1] | 3061.9 [998.4 to 7450] | 3001 [1056 to 7034.8] | 3151.2 [1003.5 to 7433.2]
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S Hexapro_293F_PPF-50-N at Month 2-Total | 1470.5 [708.7 to 3436.8] | 1275.8 [704.8 to 2869.2] | 1574.2 [704.8 to 3598.8] | 1739.8 [679 to 3617.2] | 1724 [691.9 to 3457.2] | 1177 [642.5 to 3266.8] | 1341.2 [663.1 to 3457.2] | 1315 [615.4 to 3061.9] | 1527.5 [698.3 to 3436.8] | 1275.8 [615.4 to 3061.9] | 1576.5 [706.1 to 3477.8]
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 0-Total | 1629.8 [297.8 to 4646.2] | 3462.6 [877.6 to 7865.3] | 739.8 [64.8 to 1493.8] | 1596 [524.1 to 3955.9] | 2043 [739.8 to 5212] | 2536.5 [906.7 to 6080.9] | 2051.2 [920.6 to 3452.1] | 5076.8 [1966.5 to 9966.8] | 2043 [975.5 to 4485.8] | 2627.8 [701.2 to 6589.3] | 2188.4 [929.8 to 5065.4]
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S Hexapro_293F_PPF-50-Y at Month 2-Total | 726.2 [195.2 to 2527.2] | 1844 [462.6 to 5081.6] | 1038.5 [129.2 to 1260.8] | 1076.5 [726.5 to 2339.8] | 1245.8 [637.8 to 2869.2] | 1578.8 [815.2 to 3598.8] | 1480.8 [710 to 2719.8] | 2486.2 [897.5 to 4301.5] | 1088.1 [270.4 to 1856.5] | 2486.2 [817.5 to 3868] | 1118 [387.4 to 2372.1]
  SARS-CoV-2 S1 C His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S1 C His-50-N at Month 0-Total | 2394.5 [651.1 to 6589.9] | 1982.5 [613.6 to 6713] | 2510.4 [747.1 to 6663.3] | 3158.4 [852.5 to 8476.1] | 2897.8 [863.5 to 7763.1] | 2319.2 [654 to 7507.2] | 2408 [637.4 to 6835.2] | 1943.6 [521.9 to 6082.2] | 2338.9 [613.3 to 6666.4] | 2299.5 [686.5 to 6668] | 2385.5 [607.8 to 6904]
  SARS-CoV-2 S1 C His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1 C His-50-N at Month 2-Total | 728.9 [281.6 to 2464.1] | 685.8 [280.2 to 1988.8] | 806.8 [282 to 2490] | 1005.5 [334.5 to 2631.8] | 806.8 [308.2 to 2512.5] | 683.2 [241.2 to 1775.4] | 806.8 [255.8 to 2389] | 685.8 [246.6 to 2256.9] | 783.6 [281.6 to 2355.8] | 683.2 [264.5 to 1775.4] | 799.8 [280.7 to 2317.3]
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S1 C His-50-Y at Month 0-Total | 1173.5 [155 to 2577.8] | 2609.4 [634.1 to 5814.9] | 398 [124 to 1588.5] | 1189 [319.9 to 3025.5] | 1594 [398 to 4820.5] | 1974.8 [592.3 to 5858.1] | 1538.5 [380.4 to 4476.8] | 4003.8 [1591.2 to 9347] | 1236.2 [721.6 to 4351.2] | 1995.5 [235.4 to 5414.5] | 1542.1 [682.1 to 4819.2]
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1 C His-50-Y at Month 2-Total | 507.4 [125.2 to 1239.4] | 1246.8 [213 to 3447.4] | 233.8 [150.1 to 742] | 639.2 [227.8 to 1860.9] | 692 [233.8 to 1988.8] | 1005.5 [308 to 2569.5] | 587 [332 to 2212] | 1988.8 [1246.8 to 4975.8] | 381.6 [187.4 to 2226.2] | 1988.8 [262.8 to 2615.5] | 605.4 [204.6 to 2168.4]
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 S1S2 ECD His-50-N at Month 0-Total | 4301.8 [1626.6 to 8135.1] | 4204.2 [1601.6 to 7936.2] | 4301.8 [1664.3 to 8056.5] | 5034.8 [1863.1 to 8639.4] | 4939.6 [1843.6 to 8625.1] | 4170.8 [1598.2 to 7188.2] | 4166.2 [1552.1 to 7669.7] | 3801.1 [1380.8 to 6992.2] | 4313.2 [1631.4 to 8081] | 3988.2 [1550.5 to 7227.2] | 4304 [1622.6 to 8008]
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 S1S2 ECD His-50-N at Month 2-Total | 3782 [1942.9 to 5202.2] | 3754.5 [1739.2 to 5279.2] | 3765.8 [1901.5 to 5176.5] | 3765.8 [1956.8 to 5881] | 3751.8 [1820.4 to 5848] | 3751.8 [1352.8 to 4472] | 3754.5 [1588.9 to 5094.6] | 3751.8 [1588.9 to 4887.4] | 3782 [1860.9 to 5202.2] | 3751.8 [1588.9 to 5094.6] | 3882.9 [1735.3 to 5135.6]
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 0-Total | 1898 [909.8 to 3229.2] | 3958.9 [1487.8 to 7725.8] | 1028.2 [186.8 to 2677.8] | 2637 [1038.6 to 5050.4] | 3327.8 [1218 to 6484.2] | 3883.9 [1519.8 to 8689.6] | 3819 [1530.1 to 8144.5] | 6570.5 [3450.2 to 12725.8] | 2637 [1110.9 to 5671.4] | 4747.5 [1559.6 to 9377.4] | 3316.1 [1332.6 to 6684.9]
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 S1S2 ECD His-50-Y at Month 2-Total | 2216.5 [439.8 to 4718] | 4113.8 [1691.4 to 5094.6] | 3754.5 [439.4 to 4698.2] | 3754.5 [1231.1 to 4699.2] | 4024.8 [1349.2 to 4994.5] | 3765.8 [2247.2 to 6445.2] | 4663.8 [2247.2 to 5881] | 5377.8 [4072.8 to 6530.8] | 3758.8 [952.9 to 5015.3] | 4072.8 [2388.8 to 5377.8] | 3625 [2041.4 to 5548.4]
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total: number analyzed (Participants) | 348 | 251 | 352 | 274 | 208 | 189 | 334 | 326 | 330 | 285 | 299
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 0-Total | 5887.6 [2353.9 to 11713.9] | 5561.2 [2254.1 to 11675.2] | 6100.2 [2466.4 to 11901.9] | 7121.5 [2726.7 to 12942.1] | 6966.2 [2841.6 to 13160.5] | 5866 [2259.5 to 11578.8] | 5874.6 [2188.8 to 11854.2] | 5140.5 [1839.7 to 11182.2] | 6004.9 [2171.1 to 11649.2] | 5596.8 [2259.5 to 11463.5] | 6126.5 [2173.5 to 11625.8]
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2 spike (PreS Nexelis)-50-N at Month 2-Total | 3073.1 [1801.4 to 6992.8] | 2872.8 [1753 to 5526.5] | 3058.8 [1753 to 7225.5] | 3528.5 [1817.5 to 7225.5] | 3087.5 [1819.5 to 6889.6] | 2834.8 [1532.9 to 7080] | 3003.2 [1637.8 to 7051.1] | 2872.8 [1382 to 6418.9] | 3031 [1732.6 to 6992.8] | 2604.8 [1499.1 to 6773] | 3073.1 [1770.1 to 7109.4]
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total: number analyzed (Participants) | 25 | 122 | 21 | 99 | 165 | 184 | 39 | 47 | 43 | 88 | 74
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 0-Total | 2540 [847.5 to 6597.5] | 5649.4 [1964.1 to 11326.7] | 1798 [257 to 3157] | 3157 [1381.9 to 6686.5] | 4603.8 [1663.5 to 9602.5] | 5388.6 [2087.1 to 11423.8] | 3981.8 [2100.6 to 7298] | 10308.2 [4789.4 to 15768] | 4522 [2228.6 to 11140] | 5840.5 [1625.8 to 12851] | 4577 [2032.5 to 11164]
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2 spike (PreS Nexelis)-50-Y at Month 2-Total | 1485.6 [625 to 3958.3] | 4067 [1010 to 8654.9] | 2278.8 [549.8 to 3108] | 2519.5 [1520.6 to 5080.2] | 2807 [1369.8 to 6934.5] | 3087.5 [1817.5 to 6611.5] | 2816.5 [2093.5 to 5510.2] | 5988.8 [2231.5 to 9204] | 2629.8 [674.5 to 4857.8] | 5119.8 [2167.2 to 7942.2] | 2399.1 [1180.8 to 5810.9]
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total: number analyzed (Participants) | 254 | 174 | 259 | 206 | 149 | 130 | 248 | 236 | 233 | 204 | 214
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 0-Total | 1744.4 [300.6 to 5873.2] | 1398.4 [216.4 to 5873.2] | 1690.8 [295.6 to 5638.1] | 2149.9 [317.8 to 7224.1] | 1948.2 [245 to 7281.8] | 1547.2 [225.1 to 5986.4] | 1646.5 [323.4 to 5370.8] | 1360.8 [224.6 to 4783.1] | 1593.5 [226 to 6049.8] | 1667.2 [323.2 to 5936.5] | 1592 [225.1 to 5443.4]
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total: number analyzed (Participants) | 92 | 73 | 93 | 65 | 51 | 55 | 87 | 91 | 92 | 75 | 86
  SARS-CoV-2-NTD-AVI Biotin-50-N at Month 2-Total | 407.9 [145.1 to 1527.6] | 342 [143.2 to 1132] | 409 [144 to 1578] | 454.2 [154 to 2098] | 443.8 [148.6 to 1727.5] | 286.8 [113.4 to 1250.8] | 406.8 [137.4 to 1450.4] | 286.8 [126.6 to 1340.5] | 385 [140.1 to 1420.2] | 311.8 [141.9 to 1373.6] | 352.6 [133.9 to 1348.9]
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total: number analyzed (Participants) | 21 | 101 | 16 | 69 | 126 | 145 | 27 | 39 | 42 | 71 | 61
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 0-Total | 359.8 [124 to 906.8] | 1740 [295.8 to 4387.5] | 390.1 [88.1 to 679] | 825 [182.2 to 1938.8] | 1306.2 [275.6 to 3696.6] | 1593.5 [284.8 to 4236.5] | 533.5 [83.1 to 3520.4] | 2728.8 [1067.5 to 8798.9] | 1297 [422.6 to 3501.1] | 1256.2 [101.8 to 3551.5] | 1329.8 [419.8 to 3966.5]
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total: number analyzed (Participants) | 8 | 27 | 7 | 35 | 49 | 45 | 13 | 9 | 8 | 25 | 14
  SARS-CoV-2-NTD-AVI Biotin-50-Y at Month 2-Total | 143.4 [71.1 to 525.2] | 532.8 [143.4 to 2287.5] | 145.5 [123.4 to 331.5] | 214.8 [135.2 to 617.4] | 283 [139.8 to 1118.8] | 552.5 [160.2 to 1510.8] | 254.5 [143.2 to 1357.2] | 1132 [443.8 to 5594.5] | 387.8 [176.7 to 1948.9] | 553 [143.2 to 1510.8] | 560.5 [197.1 to 1606]

52. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Comorbidity Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: COPD/Asthma/Emphysema
- Group 2: Diabetes
- Group 3: HIV/AIDS
- Group 4: Hypertension
- Group 5: Smoking Ever
- Group 6: Smoking Now
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388
Participants
  VRC7480_G614-N at Month 0-Total: number analyzed (Participants) | 332 | 324 | 328 | 283 | 207 | 331
  VRC7480_G614-N at Month 0-Total | 301 | 292 | 296 | 265 | 191 | 303
  VRC7480_G614-N at Month 12-Total: number analyzed (Participants) | 19 | 20 | 0 | 16 | 6 | 15
  VRC7480_G614-N at Month 12-Total | 18 | 20 |  | 15 | 6 | 15
  VRC7480_G614-N at Month 2-Total: number analyzed (Participants) | 193 | 196 | 188 | 164 | 120 | 191
  VRC7480_G614-N at Month 2-Total | 171 | 171 | 165 | 149 | 106 | 168
  VRC7480_G614-N at Month 4-Total: number analyzed (Participants) | 21 | 21 | 0 | 16 | 10 | 17
  VRC7480_G614-N at Month 4-Total | 20 | 19 |  | 15 | 10 | 17
  VRC7480_G614-Y at Month 0-Total: number analyzed (Participants) | 39 | 47 | 43 | 88 | 164 | 40
  VRC7480_G614-Y at Month 0-Total | 34 | 43 | 39 | 70 | 144 | 32
  VRC7480_G614-Y at Month 12-Total: number analyzed (Participants) | 4 | 3 | 23 | 7 | 17 | 8
  VRC7480_G614-Y at Month 12-Total | 4 | 2 | 22 | 7 | 16 | 7
  VRC7480_G614-Y at Month 2-Total: number analyzed (Participants) | 23 | 20 | 28 | 52 | 96 | 25
  VRC7480_G614-Y at Month 2-Total | 20 | 20 | 26 | 42 | 85 | 23
  VRC7480_G614-Y at Month 4-Total: number analyzed (Participants) | 3 | 3 | 24 | 8 | 14 | 7
  VRC7480_G614-Y at Month 4-Total | 2 | 3 | 22 | 7 | 12 | 5

53. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Comorbidity Group Among America Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2,3,4, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388
Titer
  VRC7480_G614-ID50-N at Month 0-Peru: number analyzed (Participants) | 168 | 159 | 162 | 152 | 125 | 170
  VRC7480_G614-ID50-N at Month 0-Peru | 968.4 [227.3 to 3639.6] | 848.1 [209.2 to 2962.4] | 994.9 [237.4 to 3617.3] | 961.9 [226.2 to 3611.1] | 983.4 [328.7 to 3161.2] | 978.7 [289.6 to 3617.3]
  VRC7480_G614-ID50-N at Month 0-Total: number analyzed (Participants) | 332 | 324 | 328 | 283 | 207 | 331
  VRC7480_G614-ID50-N at Month 0-Total | 493.3 [93.3 to 1874.2] | 367.1 [84.5 to 1654.7] | 475.2 [93.3 to 1874.2] | 410.6 [101.7 to 1836.3] | 618.6 [144.1 to 1912.1] | 522.1 [109.5 to 1939.2]
  VRC7480_G614-ID50-N at Month 0-USA: number analyzed (Participants) | 164 | 165 | 166 | 131 | 82 | 161
  VRC7480_G614-ID50-N at Month 0-USA | 241.8 [52.1 to 769.5] | 190.8 [52.8 to 603.2] | 238.8 [53.1 to 714.8] | 190.8 [58.7 to 553.1] | 226.3 [62 to 627.5] | 256.5 [67.7 to 749]
  VRC7480_G614-ID50-N at Month 12-Peru: number analyzed (Participants) | 7 | 7 | 0 | 7 | 4 | 7
  VRC7480_G614-ID50-N at Month 12-Peru | 289.6 [92.7 to 678.9] | 289.6 [92.7 to 678.9] |  | 289.6 [92.7 to 678.9] | 92.70 [55.9 to 212.9] | 289.6 [92.7 to 678.9]
  VRC7480_G614-ID50-N at Month 12-Total: number analyzed (Participants) | 19 | 20 | 0 | 16 | 6 | 15
  VRC7480_G614-ID50-N at Month 12-Total | 281.8 [89.2 to 549.9] | 318.0 [108.5 to 633.4] |  | 204.9 [63.9 to 445.6] | 91.50 [61.5 to 119.6] | 245.7 [115.5 to 460.7]
  VRC7480_G614-ID50-N at Month 12-USA: number analyzed (Participants) | 12 | 13 | 0 | 9 | 2 | 8
  VRC7480_G614-ID50-N at Month 12-USA | 263.8 [99.9 to 475] | 346.4 [113.2 to 608.8] |  | 117.8 [60.3 to 411.9] | 89.00 [74.6 to 103.4] | 239.0 [116.6 to 367.4]
  VRC7480_G614-ID50-N at Month 2-Peru: number analyzed (Participants) | 100 | 95 | 95 | 92 | 75 | 100
  VRC7480_G614-ID50-N at Month 2-Peru | 196.3 [46.8 to 558.9] | 152.2 [40.6 to 351.6] | 152.2 [43.4 to 420.5] | 186.6 [46.8 to 464.3] | 213.0 [53.3 to 572.9] | 196.3 [47.4 to 504.5]
  VRC7480_G614-ID50-N at Month 2-Total: number analyzed (Participants) | 193 | 196 | 188 | 164 | 120 | 191
  VRC7480_G614-ID50-N at Month 2-Total | 134.2 [39.1 to 430.5] | 105.1 [37.4 to 343.5] | 105.1 [38.7 to 349.1] | 96.20 [39.7 to 343.5] | 160.2 [47.4 to 461.4] | 134.2 [42.3 to 416.7]
  VRC7480_G614-ID50-N at Month 2-USA: number analyzed (Participants) | 93 | 101 | 93 | 72 | 45 | 91
  VRC7480_G614-ID50-N at Month 2-USA | 88.30 [35.4 to 318.9] | 88.30 [35.4 to 282.8] | 88.30 [35.4 to 325.7] | 59.40 [36.6 to 206] | 88.30 [39.1 to 237] | 91.20 [38.3 to 333.7]
  VRC7480_G614-ID50-N at Month 4-Peru: number analyzed (Participants) | 9 | 9 | 0 | 9 | 6 | 9
  VRC7480_G614-ID50-N at Month 4-Peru | 151.7 [84.8 to 245.7] | 151.7 [84.8 to 245.7] |  | 151.7 [84.8 to 245.7] | 239.0 [142.9 to 370.4] | 151.7 [84.8 to 245.7]
  VRC7480_G614-ID50-N at Month 4-Total: number analyzed (Participants) | 21 | 21 | 0 | 16 | 10 | 17
  VRC7480_G614-ID50-N at Month 4-Total | 232.2 [113.2 to 411.9] | 187.1 [94.3 to 411.9] |  | 169.4 [78.6 to 293] | 239.0 [137 to 440.6] | 245.7 [120.2 to 411.9]
  VRC7480_G614-ID50-N at Month 4-USA: number analyzed (Participants) | 12 | 12 | 0 | 7 | 4 | 8
  VRC7480_G614-ID50-N at Month 4-USA | 267.6 [119.6 to 448.2] | 220.2 [111.9 to 448.2] |  | 187.1 [89.6 to 350.5] | 318.6 [170.4 to 517.4] | 314.1 [236.8 to 517.4]
  VRC7480_G614-ID50-Y at Month 0-Peru: number analyzed (Participants) | 9 | 18 | 15 | 25 | 52 | 7
  VRC7480_G614-ID50-Y at Month 0-Peru | 822.9 [332 to 1611] | 3196 [1616.4 to 7903.4] | 522.1 [276.9 to 1267.3] | 1141 [441.7 to 3161.2] | 609.9 [184.7 to 3745.2] | 197.1 [76.2 to 438.7]
  VRC7480_G614-ID50-Y at Month 0-Total: number analyzed (Participants) | 39 | 47 | 43 | 88 | 164 | 40
  VRC7480_G614-ID50-Y at Month 0-Total | 216.0 [81.6 to 1289.4] | 1196 [495.3 to 3195.5] | 347.6 [86.5 to 1125.9] | 594.9 [48 to 1590.3] | 336.8 [67.2 to 1617.1] | 125.6 [10 to 723.6]
  VRC7480_G614-ID50-Y at Month 0-USA: number analyzed (Participants) | 30 | 29 | 28 | 63 | 112 | 33
  VRC7480_G614-ID50-Y at Month 0-USA | 197.2 [80.5 to 642.4] | 608.3 [216 to 1333.7] | 169.2 [64.6 to 1072.5] | 462.9 [21.3 to 1214.1] | 238.9 [51.3 to 985.2] | 121.1 [10 to 740]
  VRC7480_G614-ID50-Y at Month 12-Peru: number analyzed (Participants) | 0 | 0 | 7 | 0 | 3 | 0
  VRC7480_G614-ID50-Y at Month 12-Peru |  |  | 289.6 [92.7 to 678.9] |  | 866.7 [578.1 to 915.5] |
  VRC7480_G614-ID50-Y at Month 12-Total: number analyzed (Participants) | 4 | 3 | 23 | 7 | 17 | 8
  VRC7480_G614-ID50-Y at Month 12-Total | 322.1 [197.8 to 485.8] | 232.2 [118.6 to 239] | 281.8 [103.8 to 549.9] | 281.8 [239 to 716.7] | 346.4 [232.2 to 707.2] | 346.9 [85.5 to 633.4]
  VRC7480_G614-ID50-Y at Month 12-USA: number analyzed (Participants) | 4 | 3 | 16 | 7 | 14 | 8
  VRC7480_G614-ID50-Y at Month 12-USA | 322.1 [197.8 to 485.8] | 232.2 [118.6 to 239] | 263.8 [108.5 to 475] | 281.8 [239 to 716.7] | 314.1 [142.9 to 564.2] | 346.9 [85.5 to 633.4]
  VRC7480_G614-ID50-Y at Month 2-Peru: number analyzed (Participants) | 6 | 11 | 11 | 14 | 31 | 6
  VRC7480_G614-ID50-Y at Month 2-Peru | 95.30 [19.9 to 131.8] | 1087 [378.9 to 1402.8] | 447.6 [186.6 to 713.1] | 198.0 [19.6 to 545.6] | 86.20 [20.3 to 334.8] | 39.90 [15.1 to 77]
  VRC7480_G614-ID50-Y at Month 2-Total: number analyzed (Participants) | 23 | 20 | 28 | 52 | 96 | 25
  VRC7480_G614-ID50-Y at Month 2-Total | 133.7 [58.9 to 310.5] | 443.2 [212.7 to 1229.1] | 201.4 [112.9 to 599.9] | 176.0 [59.5 to 578.9] | 96.20 [30.3 to 341.9] | 122.3 [30.6 to 253.3]
  VRC7480_G614-ID50-Y at Month 2-USA: number analyzed (Participants) | 17 | 9 | 17 | 38 | 65 | 19
  VRC7480_G614-ID50-Y at Month 2-USA | 157.2 [84.8 to 355.4] | 318.9 [211.7 to 341.6] | 157.2 [84.8 to 430.5] | 167.0 [85.6 to 562.1] | 125.4 [37 to 337.1] | 157.2 [41.9 to 295.2]
  VRC7480_G614-ID50-Y at Month 4-Peru: number analyzed (Participants) | 0 | 0 | 9 | 0 | 3 | 0
  VRC7480_G614-ID50-Y at Month 4-Peru |  |  | 151.7 [84.8 to 245.7] |  | 60.30 [44.8 to 106] |
  VRC7480_G614-ID50-Y at Month 4-Total: number analyzed (Participants) | 3 | 3 | 24 | 8 | 14 | 7
  VRC7480_G614-ID50-Y at Month 4-Total | 94.30 [49.7 to 410.3] | 281.8 [170.4 to 500.4] | 209.7 [91.9 to 420.9] | 314.1 [111.9 to 517.4] | 134.7 [59.3 to 330.2] | 94.30 [32 to 282.7]
  VRC7480_G614-ID50-Y at Month 4-USA: number analyzed (Participants) | 3 | 3 | 15 | 8 | 11 | 7
  VRC7480_G614-ID50-Y at Month 4-USA | 94.30 [49.7 to 410.3] | 281.8 [170.4 to 500.4] | 253.3 [106.1 to 448.9] | 314.1 [111.9 to 517.4] | 253.3 [76.6 to 397] | 94.30 [32 to 282.7]
  VRC7480_G614-ID80-N at Month 0-Peru: number analyzed (Participants) | 168 | 159 | 162 | 152 | 125 | 170
  VRC7480_G614-ID80-N at Month 0-Peru | 214.7 [57.9 to 685.8] | 183.0 [55.4 to 603.6] | 222.7 [60.8 to 679.1] | 211.1 [57.9 to 631.9] | 225.3 [80.4 to 644.9] | 222.7 [74.9 to 679.1]
  VRC7480_G614-ID80-N at Month 0-Total: number analyzed (Participants) | 332 | 324 | 328 | 283 | 207 | 331
  VRC7480_G614-ID80-N at Month 0-Total | 126.4 [30.3 to 420.2] | 104.4 [27.9 to 365.4] | 126.1 [30.1 to 507.3] | 107.9 [31 to 403.7] | 147.1 [37.8 to 527.8] | 133.2 [32.2 to 527.8]
  VRC7480_G614-ID80-N at Month 0-USA: number analyzed (Participants) | 164 | 165 | 166 | 131 | 82 | 161
  VRC7480_G614-ID80-N at Month 0-USA | 56.00 [19.8 to 171.1] | 48.00 [18.7 to 146] | 55.20 [21.1 to 163.3] | 48.00 [21.5 to 145] | 52.00 [22.3 to 151.8] | 67.00 [22.8 to 171.1]
  VRC7480_G614-ID80-N at Month 12-Peru: number analyzed (Participants) | 7 | 7 | 0 | 7 | 4 | 7
  VRC7480_G614-ID80-N at Month 12-Peru | 104.3 [46.4 to 197.3] | 104.3 [46.4 to 197.3] |  | 104.3 [46.4 to 197.3] | 46.40 [36.4 to 68.8] | 104.3 [46.4 to 197.3]
  VRC7480_G614-ID80-N at Month 12-Total: number analyzed (Participants) | 19 | 20 | 0 | 16 | 6 | 15
  VRC7480_G614-ID80-N at Month 12-Total | 104.3 [40.7 to 158.8] | 116.0 [42.4 to 183.1] |  | 75.50 [29.1 to 141.2] | 45.10 [16.6 to 46.5] | 87.30 [45.1 to 131.8]
  VRC7480_G614-ID80-N at Month 12-USA: number analyzed (Participants) | 12 | 13 | 0 | 9 | 2 | 8
  VRC7480_G614-ID80-N at Month 12-USA | 92.50 [34 to 141.8] | 120.4 [37.3 to 182.2] |  | 44.10 [24.4 to 128.3] | 25.80 [16.6 to 34.9] | 80.40 [42.4 to 122.4]
  VRC7480_G614-ID80-N at Month 2-Peru: number analyzed (Participants) | 100 | 95 | 95 | 92 | 75 | 100
  VRC7480_G614-ID80-N at Month 2-Peru | 57.40 [20.8 to 157.1] | 39.80 [10 to 131.7] | 39.80 [15.2 to 145.6] | 54.60 [20.8 to 145.9] | 65.00 [25.9 to 161.2] | 57.40 [22.5 to 148.2]
  VRC7480_G614-ID80-N at Month 2-Total: number analyzed (Participants) | 193 | 196 | 188 | 164 | 120 | 191
  VRC7480_G614-ID80-N at Month 2-Total | 38.60 [10 to 137.3] | 35.40 [10 to 120.5] | 35.50 [10 to 122.4] | 33.50 [10 to 118.5] | 41.60 [10 to 145.9] | 38.40 [10 to 139.5]
  VRC7480_G614-ID80-N at Month 2-USA: number analyzed (Participants) | 93 | 101 | 93 | 72 | 45 | 91
  VRC7480_G614-ID80-N at Month 2-USA | 30.00 [10 to 67.1] | 30.00 [10 to 80.6] | 30.00 [10 to 67.1] | 22.80 [10 to 53.1] | 30.00 [10 to 51.6] | 31.40 [10 to 79.1]
  VRC7480_G614-ID80-N at Month 4-Peru: number analyzed (Participants) | 9 | 9 | 0 | 9 | 6 | 9
  VRC7480_G614-ID80-N at Month 4-Peru | 55.70 [30.6 to 87.3] | 55.70 [30.6 to 87.3] |  | 55.70 [30.6 to 87.3] | 80.40 [46.3 to 140.7] | 55.70 [30.6 to 87.3]
  VRC7480_G614-ID80-N at Month 4-Total: number analyzed (Participants) | 21 | 21 | 0 | 16 | 10 | 17
  VRC7480_G614-ID80-N at Month 4-Total | 73.50 [37.3 to 127.8] | 62.60 [30.6 to 127.8] |  | 59.20 [29.1 to 97.4] | 80.40 [50.6 to 153.4] | 80.70 [46.6 to 138.2]
  VRC7480_G614-ID80-N at Month 4-USA: number analyzed (Participants) | 12 | 12 | 0 | 7 | 4 | 8
  VRC7480_G614-ID80-N at Month 4-USA | 96.10 [46 to 130.4] | 71.70 [40.7 to 130.4] |  | 62.60 [35.5 to 104.2] | 100.4 [58.6 to 147.9] | 116.0 [76.2 to 147.9]
  VRC7480_G614-ID80-Y at Month 0-Peru: number analyzed (Participants) | 9 | 18 | 15 | 25 | 52 | 7
  VRC7480_G614-ID80-Y at Month 0-Peru | 209.0 [100.9 to 354.6] | 739.4 [278.5 to 1080.6] | 147.1 [67.7 to 259.1] | 354.1 [102.9 to 695.5] | 143.2 [47.1 to 748.7] | 54.70 [25.6 to 106.1]
  VRC7480_G614-ID80-Y at Month 0-Total: number analyzed (Participants) | 39 | 47 | 43 | 88 | 164 | 40
  VRC7480_G614-ID80-Y at Month 0-Total | 83.90 [26.1 to 259.8] | 222.3 [128.8 to 658.5] | 81.50 [25.2 to 259.1] | 143.9 [11.3 to 400.1] | 104.4 [22.7 to 287.5] | 34.60 [10 to 142.6]
  VRC7480_G614-ID80-Y at Month 0-USA: number analyzed (Participants) | 30 | 29 | 28 | 63 | 112 | 33
  VRC7480_G614-ID80-Y at Month 0-USA | 54.00 [25.2 to 165.3] | 164.6 [54.5 to 260.5] | 52.40 [18.6 to 246.4] | 126.6 [10 to 243.2] | 75.30 [16.9 to 211.6] | 32.50 [10 to 144]
  VRC7480_G614-ID80-Y at Month 12-Peru: number analyzed (Participants) | 0 | 0 | 7 | 0 | 3 | 0
  VRC7480_G614-ID80-Y at Month 12-Peru |  |  | 104.3 [46.4 to 197.3] |  | 259.2 [181.7 to 323.3] |
  VRC7480_G614-ID80-Y at Month 12-Total: number analyzed (Participants) | 4 | 3 | 23 | 7 | 17 | 8
  VRC7480_G614-ID80-Y at Month 12-Total | 122.9 [73.2 to 166.2] | 73.50 [39.2 to 80.4] | 104.3 [40.7 to 170.4] | 111.5 [80.4 to 187.6] | 120.4 [73.5 to 185.8] | 135.0 [29.1 to 184]
  VRC7480_G614-ID80-Y at Month 12-USA: number analyzed (Participants) | 4 | 3 | 16 | 7 | 14 | 8
  VRC7480_G614-ID80-Y at Month 12-USA | 122.9 [73.2 to 166.2] | 73.50 [39.2 to 80.4] | 99.40 [35.6 to 164.4] | 111.5 [80.4 to 187.6] | 116.0 [46.3 to 176.3] | 135.0 [29.1 to 184]
  VRC7480_G614-ID80-Y at Month 2-Peru: number analyzed (Participants) | 6 | 11 | 11 | 14 | 31 | 6
  VRC7480_G614-ID80-Y at Month 2-Peru | 31.50 [9.9 to 39.1] | 311.5 [117 to 462] | 127.8 [63.8 to 183.2] | 58.60 [10.9 to 162.3] | 26.60 [10 to 115.6] | 15.50 [10 to 31.5]
  VRC7480_G614-ID80-Y at Month 2-Total: number analyzed (Participants) | 23 | 20 | 28 | 52 | 96 | 25
  VRC7480_G614-ID80-Y at Month 2-Total | 38.40 [23.4 to 95.1] | 112.0 [56.4 to 314.9] | 70.80 [41.8 to 154] | 52.60 [26.5 to 170.5] | 34.80 [10 to 105.5] | 47.60 [10 to 76.5]
  VRC7480_G614-ID80-Y at Month 2-USA: number analyzed (Participants) | 17 | 9 | 17 | 38 | 65 | 19
  VRC7480_G614-ID80-Y at Month 2-USA | 49.30 [30.6 to 156.1] | 58.80 [54.1 to 77.7] | 55.70 [30.6 to 128.3] | 52.60 [31 to 172.2] | 38.60 [10 to 80.7] | 49.90 [11.9 to 78.6]
  VRC7480_G614-ID80-Y at Month 4-Peru: number analyzed (Participants) | 0 | 0 | 9 | 0 | 3 | 0
  VRC7480_G614-ID80-Y at Month 4-Peru |  |  | 55.70 [30.6 to 87.3] |  | 13.70 [10.6 to 34.7] |
  VRC7480_G614-ID80-Y at Month 4-Total: number analyzed (Participants) | 3 | 3 | 24 | 8 | 14 | 7
  VRC7480_G614-ID80-Y at Month 4-Total | 30.60 [17.8 to 108.2] | 111.5 [67.9 to 144.2] | 68.10 [30.6 to 130.4] | 116.0 [40.7 to 147.9] | 49.90 [16.4 to 118.2] | 30.60 [14.7 to 85.9]
  VRC7480_G614-ID80-Y at Month 4-USA: number analyzed (Participants) | 3 | 3 | 15 | 8 | 11 | 7
  VRC7480_G614-ID80-Y at Month 4-USA | 30.60 [17.8 to 108.2] | 111.5 [67.9 to 144.2] | 80.70 [37.4 to 133] | 116.0 [40.7 to 147.9] | 80.70 [27.5 to 124.1] | 30.60 [14.7 to 85.9]

54. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (Nab) by Region and Comorbidity Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and comorbidity group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 372 | 372 | 372 | 372 | 372 | 372
Participants
  SARS-Cov-2 D614G-N at Month 0-Total: number analyzed (Participants) | 307 | 277 | 284 | 246 | 261 | 292
  SARS-Cov-2 D614G-N at Month 0-Total | 277 | 248 | 255 | 218 | 239 | 264
  SARS-Cov-2 D614G-N at Month 12-Total: number analyzed (Participants) | 174 | 160 | 157 | 145 | 144 | 164
  SARS-Cov-2 D614G-N at Month 12-Total | 169 | 155 | 153 | 141 | 142 | 160
  SARS-Cov-2 D614G-N at Month 2-Total: number analyzed (Participants) | 226 | 207 | 208 | 178 | 184 | 211
  SARS-Cov-2 D614G-N at Month 2-Total | 202 | 183 | 184 | 158 | 168 | 190
  SARS-Cov-2 D614G-N at Month 4-Total: number analyzed (Participants) | 219 | 197 | 200 | 174 | 178 | 200
  SARS-Cov-2 D614G-N at Month 4-Total | 200 | 178 | 182 | 158 | 168 | 186
  SARS-Cov-2 D614G-Y at Month 0-Total: number analyzed (Participants) | 16 | 46 | 39 | 77 | 62 | 31
  SARS-Cov-2 D614G-Y at Month 0-Total | 15 | 44 | 37 | 74 | 53 | 28
  SARS-Cov-2 D614G-Y at Month 12-Total: number analyzed (Participants) | 7 | 21 | 24 | 36 | 37 | 17
  SARS-Cov-2 D614G-Y at Month 12-Total | 7 | 21 | 23 | 35 | 34 | 16
  SARS-Cov-2 D614G-Y at Month 2-Total: number analyzed (Participants) | 11 | 30 | 29 | 59 | 53 | 26
  SARS-Cov-2 D614G-Y at Month 2-Total | 10 | 29 | 28 | 54 | 44 | 22
  SARS-Cov-2 D614G-Y at Month 4-Total: number analyzed (Participants) | 9 | 31 | 28 | 54 | 50 | 28
  SARS-Cov-2 D614G-Y at Month 4-Total | 8 | 30 | 26 | 50 | 40 | 22

55. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (Nab) by Region and Comorbidity Group Among Africa Cohort
Description: Neutralizing antibodies against SARS coronaviruses are measured in 293T/ACE2 cells for all HIV negative samples. MPI (maximum percent inhibition) is also measured. Positivity calls are an ID50/ID80 (50% and 80% inhibitory dose) value either >20 (the lower limit of detection (LLOD) of the assay) or MPI is between 10%-50%. The neutralizing antibody ID50/ID80 of all HIV positive samples are measured by a different assay, VSV pseudovirus neutralization assay. Positivity calls are based on whether or not any neutralization is observed through entire titration (starting dilution 1:20) with MPI between 10%-50%. For the positive calls but the neutralization does not reach 50% or 80%, ID50/ID80 titer is first estimated by Prism.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by neutralizing antibody assay (NAb) at Visit 1, 2, 3, 4, overall and by region and comorbidity group among Africa Cohort
Time Frame: Measured at Months 0, 2, 4, 12
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 372 | 372 | 372 | 372 | 372 | 372
Titer
  SARS-Cov-2 D614G-ID50-N at Month 0-RSA: number analyzed (Participants) | 225 | 201 | 207 | 180 | 186 | 210
  SARS-Cov-2 D614G-ID50-N at Month 0-RSA | 320.3 [122.8 to 1294.1] | 271.3 [86.3 to 994] | 366.3 [144.7 to 1459.7] | 278.1 [79 to 1150.1] | 416.9 [157.5 to 1624.2] | 362.2 [142.2 to 1463.4]
  SARS-Cov-2 D614G-ID50-N at Month 0-Total: number analyzed (Participants) | 307 | 277 | 284 | 246 | 261 | 292
  SARS-Cov-2 D614G-ID50-N at Month 0-Total | 309.6 [82.4 to 1298.5] | 253.5 [72.1 to 939.4] | 361.7 [113.6 to 1442.8] | 250.5 [68.6 to 1023.9] | 366.3 [126.2 to 1540.7] | 351.6 [110.3 to 1442.8]
  SARS-Cov-2 D614G-ID50-N at Month 0-non-RSA: number analyzed (Participants) | 82 | 76 | 77 | 66 | 75 | 82
  SARS-Cov-2 D614G-ID50-N at Month 0-non-RSA | 232.5 [19.3 to 1265.1] | 221.6 [10 to 677.6] | 329.4 [48.6 to 1149] | 202.8 [10 to 645.7] | 329.4 [58.3 to 1316.1] | 276 [47.5 to 1265.1]
  SARS-Cov-2 D614G-ID50-N at Month 12-RSA: number analyzed (Participants) | 106 | 98 | 93 | 88 | 83 | 96
  SARS-Cov-2 D614G-ID50-N at Month 12-RSA | 1742.4 [292.3 to 8145] | 1425.4 [256.7 to 7759.7] | 1582.1 [284.9 to 8241.1] | 1496.8 [275.5 to 7565.8] | 2820.3 [477.3 to 10782] | 2369.6 [334.5 to 9595]
  SARS-Cov-2 D614G-ID50-N at Month 12-Total: number analyzed (Participants) | 174 | 160 | 157 | 145 | 144 | 164
  SARS-Cov-2 D614G-ID50-N at Month 12-Total | 1254.7 [286.6 to 7080.4] | 848.1 [261 to 6522.5] | 830.5 [284.9 to 7123.1] | 830.5 [247.3 to 6188.3] | 1755.3 [358.2 to 7816.6] | 1577.6 [295.9 to 7302.1]
  SARS-Cov-2 D614G-ID50-N at Month 12-non-RSA: number analyzed (Participants) | 68 | 62 | 64 | 57 | 61 | 68
  SARS-Cov-2 D614G-ID50-N at Month 12-non-RSA | 636.2 [260.7 to 3480.7] | 636.2 [270.9 to 3186.7] | 636.2 [281.6 to 3957.2] | 602.8 [246.1 to 2443.4] | 702.3 [293.3 to 4599.5] | 681.2 [281.6 to 3957.2]
  SARS-Cov-2 D614G-ID50-N at Month 2-RSA: number analyzed (Participants) | 149 | 136 | 137 | 116 | 114 | 134
  SARS-Cov-2 D614G-ID50-N at Month 2-RSA | 191.6 [58.8 to 664.2] | 148.1 [57.1 to 521.1] | 198.4 [64.9 to 664.2] | 123.7 [55.4 to 508.1] | 246.2 [68.4 to 826.6] | 208 [67.1 to 780]
  SARS-Cov-2 D614G-ID50-N at Month 2-Total: number analyzed (Participants) | 226 | 207 | 208 | 178 | 184 | 211
  SARS-Cov-2 D614G-ID50-N at Month 2-Total | 147.6 [46 to 467.2] | 116.2 [40.9 to 414.5] | 155.3 [48.9 to 464.8] | 99.6 [37 to 351.8] | 155.3 [52.7 to 538.4] | 150.5 [51.7 to 514]
  SARS-Cov-2 D614G-ID50-N at Month 2-non-RSA: number analyzed (Participants) | 77 | 71 | 71 | 62 | 70 | 77
  SARS-Cov-2 D614G-ID50-N at Month 2-non-RSA | 63 [10 to 257] | 56.2 [9.1 to 237.2] | 71.4 [10 to 254.9] | 53.3 [10 to 227.5] | 80 [10 to 251.2] | 63 [10 to 252.7]
  SARS-Cov-2 D614G-ID50-N at Month 4-RSA: number analyzed (Participants) | 150 | 134 | 136 | 119 | 115 | 131
  SARS-Cov-2 D614G-ID50-N at Month 4-RSA | 310.6 [81 to 912.4] | 275.1 [75.6 to 904.8] | 337.3 [90.3 to 1237.2] | 292.5 [77.1 to 880.5] | 446.4 [108.6 to 1341.2] | 356.5 [103.6 to 1293.5]
  SARS-Cov-2 D614G-ID50-N at Month 4-Total: number analyzed (Participants) | 219 | 197 | 200 | 174 | 178 | 200
  SARS-Cov-2 D614G-ID50-N at Month 4-Total | 259.4 [75.8 to 881.9] | 235 [71.4 to 749.8] | 280.8 [87.7 to 938] | 236.8 [72.1 to 722.4] | 299.8 [94 to 1121.2] | 276.1 [87.7 to 994.3]
  SARS-Cov-2 D614G-ID50-N at Month 4-non-RSA: number analyzed (Participants) | 69 | 63 | 64 | 55 | 63 | 69
  SARS-Cov-2 D614G-ID50-N at Month 4-non-RSA | 185.4 [63.8 to 580.8] | 163 [60.4 to 528.8] | 214.4 [85.1 to 563.2] | 163 [60.4 to 465.9] | 188.7 [75.4 to 569.1] | 188.7 [71.4 to 580.8]
  SARS-Cov-2 D614G-ID50-Y at Month 0-RSA: number analyzed (Participants) | 14 | 38 | 32 | 59 | 53 | 29
  SARS-Cov-2 D614G-ID50-Y at Month 0-RSA | 361.8 [202.4 to 1767.7] | 1106.8 [488.7 to 2381] | 174.8 [59.9 to 504.2] | 689.3 [203.1 to 1606.2] | 227.1 [35.9 to 569.9] | 186.1 [26.2 to 474.5]
  SARS-Cov-2 D614G-ID50-Y at Month 0-Total: number analyzed (Participants) | 16 | 46 | 39 | 77 | 62 | 31
  SARS-Cov-2 D614G-ID50-Y at Month 0-Total | 394.8 [207 to 1402.2] | 1145.5 [488.7 to 2381] | 154.5 [52.9 to 506.9] | 689.3 [200 to 1644.9] | 199.3 [27.4 to 539.5] | 186.1 [25.7 to 435.8]
  SARS-Cov-2 D614G-ID50-Y at Month 0-non-RSA: number analyzed (Participants) | 2 | 8 | 7 | 18 | 9 | 2
  SARS-Cov-2 D614G-ID50-Y at Month 0-non-RSA | 507.9 [443 to 572.9] | 1632.8 [718.6 to 2125.5] | 103.7 [8.2 to 731.7] | 705.7 [133.1 to 1806.3] | 10 [5 to 338.1] | 174.1 [92 to 256.1]
  SARS-Cov-2 D614G-ID50-Y at Month 12-RSA: number analyzed (Participants) | 6 | 14 | 19 | 24 | 29 | 16
  SARS-Cov-2 D614G-ID50-Y at Month 12-RSA | 1246.4 [224.8 to 12091.3] | 6407.6 [1692.3 to 10890.6] | 2629.1 [1161.5 to 8464.3] | 5164.1 [361.6 to 17312.4] | 284.9 [102.7 to 1573.2] | 396.8 [93.8 to 2533.5]
  SARS-Cov-2 D614G-ID50-Y at Month 12-Total: number analyzed (Participants) | 7 | 21 | 24 | 36 | 37 | 17
  SARS-Cov-2 D614G-ID50-Y at Month 12-Total | 2196 [248.8 to 12252.1] | 3743.2 [872 to 11384.1] | 2598.1 [1007.8 to 7966.6] | 4233.8 [361.6 to 16089.4] | 247.3 [89 to 1689.3] | 246.3 [67 to 1315.3]
  SARS-Cov-2 D614G-ID50-Y at Month 12-non-RSA: number analyzed (Participants) | 1 | 7 | 5 | 12 | 8 | 1
  SARS-Cov-2 D614G-ID50-Y at Month 12-non-RSA | 9114.5 [9114.5 to 9114.5] | 872 [317.7 to 10965.7] | 2567.1 [111.6 to 3393.2] | 3155.1 [516.8 to 10496.6] | 237.5 [55.5 to 2202.8] | 10 [10 to 10]
  SARS-Cov-2 D614G-ID50-Y at Month 2-RSA: number analyzed (Participants) | 9 | 22 | 21 | 42 | 44 | 24
  SARS-Cov-2 D614G-ID50-Y at Month 2-RSA | 161.7 [93.6 to 422] | 424.4 [168 to 962.5] | 93.6 [51 to 502.2] | 308 [115.1 to 916.6] | 134.2 [10 to 271.6] | 72.9 [10 to 271.6]
  SARS-Cov-2 D614G-ID50-Y at Month 2-Total: number analyzed (Participants) | 11 | 30 | 29 | 59 | 53 | 26
  SARS-Cov-2 D614G-ID50-Y at Month 2-Total | 129.6 [78.3 to 317.6] | 424.4 [168 to 1097.9] | 66 [44.7 to 502.2] | 307 [97 to 878.3] | 120.8 [10 to 275.6] | 72.9 [10 to 274.3]
  SARS-Cov-2 D614G-ID50-Y at Month 2-non-RSA: number analyzed (Participants) | 2 | 8 | 8 | 17 | 9 | 2
  SARS-Cov-2 D614G-ID50-Y at Month 2-non-RSA | 92 [73.2 to 110.8] | 552.1 [183 to 1563.3] | 52.9 [8.2 to 217.6] | 211.4 [56.2 to 822.6] | 48.9 [5 to 337.9] | 243.5 [124.3 to 362.8]
  SARS-Cov-2 D614G-ID50-Y at Month 4-RSA: number analyzed (Participants) | 7 | 23 | 21 | 38 | 42 | 26
  SARS-Cov-2 D614G-ID50-Y at Month 4-RSA | 546.3 [286.9 to 1239.8] | 657.1 [253.4 to 1347.8] | 146.1 [66.6 to 705.2] | 528.4 [178.2 to 1415.1] | 165.5 [13.5 to 467.2] | 104.4 [10 to 467.2]
  SARS-Cov-2 D614G-ID50-Y at Month 4-Total: number analyzed (Participants) | 9 | 31 | 28 | 54 | 50 | 28
  SARS-Cov-2 D614G-ID50-Y at Month 4-Total | 474.5 [267.3 to 891.8] | 657.1 [253.4 to 1347.8] | 104.4 [54.2 to 705.4] | 528.4 [144.2 to 1382.3] | 165.5 [13.5 to 467.2] | 104.4 [10 to 452.4]
  SARS-Cov-2 D614G-ID50-Y at Month 4-non-RSA: number analyzed (Participants) | 2 | 8 | 7 | 16 | 8 | 2
  SARS-Cov-2 D614G-ID50-Y at Month 4-non-RSA | 310.4 [288.9 to 332] | 767.5 [258.2 to 1314] | 25.8 [8.2 to 598.7] | 445.3 [117.7 to 1170.2] | 145.6 [45.3 to 665.1] | 171.6 [90.8 to 252.4]
  SARS-Cov-2 D614G-ID80-N at Month 0-RSA: number analyzed (Participants) | 225 | 201 | 207 | 180 | 186 | 210
  SARS-Cov-2 D614G-ID80-N at Month 0-RSA | 82.2 [34.2 to 294.2] | 62.8 [30.9 to 210.9] | 100.1 [35.2 to 357] | 61.3 [26.6 to 238.2] | 100.5 [37.1 to 398.2] | 98.2 [35.1 to 357.8]
  SARS-Cov-2 D614G-ID80-N at Month 0-Total: number analyzed (Participants) | 307 | 277 | 284 | 246 | 261 | 292
  SARS-Cov-2 D614G-ID80-N at Month 0-Total | 79.4 [29 to 276.7] | 58.2 [24.6 to 207.6] | 98.5 [32 to 322.8] | 55.1 [24.4 to 222.7] | 100.1 [34.3 to 355.6] | 93 [31.7 to 332]
  SARS-Cov-2 D614G-ID80-N at Month 0-non-RSA: number analyzed (Participants) | 82 | 76 | 77 | 66 | 75 | 82
  SARS-Cov-2 D614G-ID80-N at Month 0-non-RSA | 47.8 [10 to 255.3] | 45.7 [10 to 184.4] | 50.4 [23.8 to 233.6] | 43.4 [10 to 181.4] | 95.8 [24.6 to 268.6] | 49.6 [13.5 to 255.3]
  SARS-Cov-2 D614G-ID80-N at Month 12-RSA: number analyzed (Participants) | 106 | 98 | 93 | 88 | 83 | 96
  SARS-Cov-2 D614G-ID80-N at Month 12-RSA | 492.2 [106.2 to 2650.7] | 345.7 [62.8 to 1910] | 392.2 [62.8 to 2760.8] | 390.9 [62.8 to 1749.9] | 794.6 [135.6 to 3207.8] | 694.3 [113.8 to 2878.6]
  SARS-Cov-2 D614G-ID80-N at Month 12-Total: number analyzed (Participants) | 174 | 160 | 157 | 145 | 144 | 164
  SARS-Cov-2 D614G-ID80-N at Month 12-Total | 295.6 [97.4 to 1735.7] | 227.3 [68.3 to 1550.2] | 224 [70.6 to 1837] | 224 [63.9 to 1357] | 508.1 [122.3 to 2347.2] | 407 [104.8 to 2126.8]
  SARS-Cov-2 D614G-ID80-N at Month 12-non-RSA: number analyzed (Participants) | 68 | 62 | 64 | 57 | 61 | 68
  SARS-Cov-2 D614G-ID80-N at Month 12-non-RSA | 179.1 [87 to 952.1] | 179.1 [94.3 to 907.5] | 179.1 [98.1 to 978.7] | 173.2 [70.6 to 757.7] | 190.8 [104.7 to 1000] | 187.5 [98.1 to 978.7]
  SARS-Cov-2 D614G-ID80-N at Month 2-RSA: number analyzed (Participants) | 149 | 136 | 137 | 116 | 114 | 134
  SARS-Cov-2 D614G-ID80-N at Month 2-RSA | 42 [13.4 to 173.5] | 39.3 [10 to 143.2] | 43.7 [20.9 to 174.8] | 37.7 [10 to 141.3] | 75.4 [22.3 to 187.2] | 61.4 [21.8 to 185.1]
  SARS-Cov-2 D614G-ID80-N at Month 2-Total: number analyzed (Participants) | 226 | 207 | 208 | 178 | 184 | 211
  SARS-Cov-2 D614G-ID80-N at Month 2-Total | 36.4 [10 to 137.2] | 34.4 [10 to 117] | 37.7 [10 to 134] | 33.5 [10 to 104.8] | 38.8 [10 to 153.6] | 37.7 [10 to 147.8]
  SARS-Cov-2 D614G-ID80-N at Month 2-non-RSA: number analyzed (Participants) | 77 | 71 | 71 | 62 | 70 | 77
  SARS-Cov-2 D614G-ID80-N at Month 2-non-RSA | 23.6 [10 to 65.5] | 22.8 [7.5 to 52] | 25.2 [10 to 59.2] | 22.6 [10 to 43.2] | 25.7 [10 to 62.4] | 24.5 [10 to 53]
  SARS-Cov-2 D614G-ID80-N at Month 4-RSA: number analyzed (Participants) | 150 | 134 | 136 | 119 | 115 | 131
  SARS-Cov-2 D614G-ID80-N at Month 4-RSA | 90.6 [27.3 to 209.3] | 83.7 [23 to 207] | 102.4 [30.5 to 265.7] | 81.9 [22.9 to 202.1] | 118.1 [34.6 to 293.6] | 113.5 [33.7 to 271.1]
  SARS-Cov-2 D614G-ID80-N at Month 4-Total: number analyzed (Participants) | 219 | 197 | 200 | 174 | 178 | 200
  SARS-Cov-2 D614G-ID80-N at Month 4-Total | 66.6 [25.3 to 206.7] | 57.1 [23.9 to 188.9] | 84.6 [28.6 to 217.9] | 55.6 [24 to 176.3] | 96.3 [31.7 to 238.1] | 86.5 [29.1 to 226.8]
  SARS-Cov-2 D614G-ID80-N at Month 4-non-RSA: number analyzed (Participants) | 69 | 63 | 64 | 55 | 63 | 69
  SARS-Cov-2 D614G-ID80-N at Month 4-non-RSA | 43.8 [24.2 to 177.1] | 43.3 [23.9 to 150.6] | 50.2 [27.5 to 174.7] | 43.3 [24.1 to 147.2] | 48.4 [24.2 to 175.5] | 45.4 [24.2 to 177.1]
  SARS-Cov-2 D614G-ID80-Y at Month 0-RSA: number analyzed (Participants) | 14 | 38 | 32 | 59 | 53 | 29
  SARS-Cov-2 D614G-ID80-Y at Month 0-RSA | 106.7 [59.1 to 383.7] | 267.9 [120.6 to 573.9] | 46.5 [15.4 to 102.7] | 181.5 [60.1 to 420.7] | 52.2 [10 to 138.1] | 49.7 [10 to 131.6]
  SARS-Cov-2 D614G-ID80-Y at Month 0-Total: number analyzed (Participants) | 16 | 46 | 39 | 77 | 62 | 31
  SARS-Cov-2 D614G-ID80-Y at Month 0-Total | 120.8 [61.3 to 267.6] | 309.3 [120.6 to 597.9] | 42.1 [11 to 104.6] | 181.5 [58 to 465.6] | 47.8 [10 to 131.4] | 49.7 [10 to 131.2]
  SARS-Cov-2 D614G-ID80-Y at Month 0-non-RSA: number analyzed (Participants) | 2 | 8 | 7 | 18 | 9 | 2
  SARS-Cov-2 D614G-ID80-Y at Month 0-non-RSA | 144.6 [133.1 to 156] | 396.2 [143.4 to 623.4] | 28.4 [7.5 to 202.6] | 174.4 [49.3 to 574.2] | 10 [5 to 31.2] | 59.7 [34.9 to 84.6]
  SARS-Cov-2 D614G-ID80-Y at Month 12-RSA: number analyzed (Participants) | 6 | 14 | 19 | 24 | 29 | 16
  SARS-Cov-2 D614G-ID80-Y at Month 12-RSA | 378.4 [57.1 to 2969.3] | 2077.3 [472.3 to 3267.6] | 576.2 [270 to 1781.6] | 1076.4 [129.1 to 4163.6] | 62.8 [35.9 to 392.2] | 88.3 [32.1 to 458.3]
  SARS-Cov-2 D614G-ID80-Y at Month 12-Total: number analyzed (Participants) | 7 | 21 | 24 | 36 | 37 | 17
  SARS-Cov-2 D614G-ID80-Y at Month 12-Total | 694.1 [59 to 3157.7] | 971.6 [238.8 to 3310.6] | 530.3 [218.2 to 1524.3] | 1022.7 [129.1 to 3560.9] | 62.8 [34 to 601.6] | 63.9 [26.2 to 301.9]
  SARS-Cov-2 D614G-ID80-Y at Month 12-non-RSA: number analyzed (Participants) | 1 | 7 | 5 | 12 | 8 | 1
  SARS-Cov-2 D614G-ID80-Y at Month 12-non-RSA | 2587.7 [2587.7 to 2587.7] | 238.8 [89.2 to 2238.4] | 484.4 [41.8 to 600.6] | 728 [145.9 to 2451.8] | 65.9 [19.8 to 694.1] | 10 [10 to 10]
  SARS-Cov-2 D614G-ID80-Y at Month 2-RSA: number analyzed (Participants) | 9 | 22 | 21 | 42 | 44 | 24
  SARS-Cov-2 D614G-ID80-Y at Month 2-RSA | 57.3 [37.4 to 105] | 142.1 [42.8 to 202.9] | 35.2 [7.5 to 137] | 109.5 [34.6 to 197.1] | 34.3 [10 to 62.9] | 26.6 [10 to 46.2]
  SARS-Cov-2 D614G-ID80-Y at Month 2-Total: number analyzed (Participants) | 11 | 30 | 29 | 59 | 53 | 26
  SARS-Cov-2 D614G-ID80-Y at Month 2-Total | 39.3 [31.3 to 87.3] | 142.1 [41.2 to 217.1] | 29.9 [7.5 to 137] | 87.1 [32.4 to 197.5] | 33.5 [10 to 60.6] | 26.6 [10 to 54.5]
  SARS-Cov-2 D614G-ID80-Y at Month 2-non-RSA: number analyzed (Participants) | 2 | 8 | 8 | 17 | 9 | 2
  SARS-Cov-2 D614G-ID80-Y at Month 2-non-RSA | 31.7 [28.5 to 35] | 146.1 [39.3 to 419.2] | 10.2 [7.5 to 72.3] | 53 [22.5 to 197.1] | 10 [5 to 51] | 43.7 [24.3 to 63]
  SARS-Cov-2 D614G-ID80-Y at Month 4-RSA: number analyzed (Participants) | 7 | 23 | 21 | 38 | 42 | 26
  SARS-Cov-2 D614G-ID80-Y at Month 4-RSA | 147.2 [88.5 to 423.7] | 169.7 [61.2 to 295.9] | 41.1 [19.2 to 169.7] | 136.3 [39.1 to 401.5] | 38.7 [10 to 139.5] | 31.3 [10 to 153.2]
  SARS-Cov-2 D614G-ID80-Y at Month 4-Total: number analyzed (Participants) | 9 | 31 | 28 | 54 | 50 | 28
  SARS-Cov-2 D614G-ID80-Y at Month 4-Total | 139.5 [52.6 to 215.9] | 177.1 [61.2 to 306.8] | 34.7 [10.5 to 169.8] | 137.9 [36.6 to 357.4] | 38.7 [10 to 139.5] | 31.3 [10 to 144]
  SARS-Cov-2 D614G-ID80-Y at Month 4-non-RSA: number analyzed (Participants) | 2 | 8 | 7 | 16 | 8 | 2
  SARS-Cov-2 D614G-ID80-Y at Month 4-non-RSA | 66.7 [59.6 to 73.7] | 205.9 [97.5 to 391.5] | 7.5 [6.7 to 156.2] | 153.5 [37 to 288.8] | 36.1 [22.3 to 179.4] | 64 [37 to 91]

56. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Rate (ADCC) by Region and Comorbidity Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Rate by antibody-dependent cellular cytotoxicity assay (ADCC) at Visit 1, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: HIV/AIDS
- Group 2: COPD/Asthma/Emphysema
- Group 3: Diabetes
- Group 5: Smoking Now
- Group 6: Smoking Ever
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388
Participants
  Bkg. Subtracted CD107A NK Cells-I-ADCC-No at Month 0-Total: number analyzed (Participants) | 215 | 232 | 218 | 183 | 225 | 145
  Bkg. Subtracted CD107A NK Cells-I-ADCC-No at Month 0-Total | 131 | 138 | 124 | 104 | 140 | 93
  Bkg. Subtracted CD107A NK Cells-I-ADCC-Yes at Month 0-Total: number analyzed (Participants) | 41 | 24 | 38 | 73 | 31 | 111
  Bkg. Subtracted CD107A NK Cells-I-ADCC-Yes at Month 0-Total | 21 | 14 | 28 | 48 | 12 | 59
  Bkg. Subtracted CD107A NK Cells-T-ADCC-No at Month 0-Total: number analyzed (Participants) | 215 | 232 | 218 | 183 | 225 | 145
  Bkg. Subtracted CD107A NK Cells-T-ADCC-No at Month 0-Total | 126 | 140 | 127 | 114 | 140 | 95
  Bkg. Subtracted CD107A NK Cells-T-ADCC-Yes at Month 0-Total: number analyzed (Participants) | 41 | 24 | 38 | 73 | 31 | 111
  Bkg. Subtracted CD107A NK Cells-T-ADCC-Yes at Month 0-Total | 27 | 13 | 26 | 39 | 13 | 58

57. Primary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (ADCC) by Region and Comorbidity Group Among America Cohort
Description: Antibody-dependent NK cell degranulation will be measured using ADCC assay at a dilution 1:500. Two readouts will be the background-subtracted % CD107A+ NK cells for the infected cells and the background-subtracted % CD107A+ NK cells for the transfected cells. The positive responses will be called if the values of background-subtracted % CD107A+ ≥ 4.07 and ≥5.27 for the infected and transfected cells, respectively. The cutoffs are determined by mean+2SD, respectively, from the SARS-CoV-2 negative controls. Percent CD107a+ NK Cells was the response magnitudes.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by antibody-dependent cellular cytotoxicity assay (ADCC) Visit 1, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: Percent CD107a+ NK Cells
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388
Percent CD107a+ NK Cells
  Bkg. Subtracted CD107A NK Cells-I-ADCC-No at Month 0-Total: number analyzed (Participants) | 215 | 232 | 218 | 183 | 225 | 145
  Bkg. Subtracted CD107A NK Cells-I-ADCC-No at Month 0-Total | 6 [1.3 to 13.8] | 6 [1.4 to 13.6] | 4.9 [1.3 to 12.5] | 5.1 [1.4 to 13.3] | 6.6 [1.8 to 14.1] | 6.6 [1.8 to 14.9]
  Bkg. Subtracted CD107A NK Cells-I-ADCC-Yes at Month 0-Total: number analyzed (Participants) | 41 | 24 | 38 | 73 | 31 | 111
  Bkg. Subtracted CD107A NK Cells-I-ADCC-Yes at Month 0-Total | 4.2 [1.6 to 12.2] | 5 [2.2 to 14.1] | 13 [3.8 to 20.8] | 7.5 [1.4 to 15.5] | 1.8 [0.1 to 6] | 4.5 [1.1 to 11.7]
  Bkg. Subtracted CD107A NK Cells-T-ADCC-No at Month 0-Total: number analyzed (Participants) | 215 | 232 | 218 | 183 | 225 | 145
  Bkg. Subtracted CD107A NK Cells-T-ADCC-No at Month 0-Total | 6.7 [2.9 to 13.1] | 6.9 [2.9 to 13.3] | 6.4 [2.9 to 13] | 8 [3.3 to 13.5] | 8 [3.2 to 13.4] | 8.6 [3.4 to 13.7]
  Bkg. Subtracted CD107A NK Cells-T-ADCC-Yes at Month 0-Total: number analyzed (Participants) | 41 | 24 | 38 | 73 | 31 | 111
  Bkg. Subtracted CD107A NK Cells-T-ADCC-Yes at Month 0-Total | 8.2 [4.1 to 12.9] | 6.1 [3.1 to 9.6] | 10 [3.4 to 15.1] | 5.9 [2.4 to 10.2] | 4.3 [0.6 to 8.2] | 5.7 [2.6 to 11.4]

58. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate (ICS) by Region and Comorbidity Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Rate by flow cytometry at Visit 1, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0
Population: American Population with positive responders (USA and Peru only), all available data at each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
Participants
  CD4+-Any COV2-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD4+-Any COV2-N at Month 0-Peru | 139 | 105 | 143 | 138 | 104 | 91 | 135 | 128 | 132 | 124 | 125
  CD4+-Any COV2-N at Month 0-Total: number analyzed (Participants) | 341 | 246 | 344 | 269 | 204 | 185 | 328 | 319 | 322 | 281 | 293
  CD4+-Any COV2-N at Month 0-Total | 263 | 189 | 261 | 209 | 160 | 138 | 245 | 236 | 242 | 212 | 217
  CD4+-Any COV2-N at Month 0-USA: number analyzed (Participants) | 172 | 122 | 168 | 102 | 81 | 72 | 161 | 161 | 161 | 129 | 139
  CD4+-Any COV2-N at Month 0-USA | 124 | 84 | 118 | 71 | 56 | 47 | 110 | 108 | 110 | 88 | 92
  CD4+-Any COV2-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD4+-Any COV2-Y at Month 0-Peru | 4 | 38 | 0 | 5 | 39 | 52 | 8 | 15 | 11 | 19 | 18
  CD4+-Any COV2-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 96 | 161 | 180 | 37 | 46 | 43 | 84 | 72
  CD4+-Any COV2-Y at Month 0-Total | 9 | 83 | 11 | 63 | 112 | 134 | 27 | 36 | 30 | 60 | 55
  CD4+-Any COV2-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 87 | 108 | 117 | 28 | 28 | 28 | 60 | 50
  CD4+-Any COV2-Y at Month 0-USA | 5 | 45 | 11 | 58 | 73 | 82 | 19 | 21 | 19 | 41 | 37
  CD4+-E M-N at Month 0-Peru: number analyzed (Participants) | 167 | 123 | 174 | 165 | 122 | 113 | 166 | 156 | 160 | 150 | 153
  CD4+-E M-N at Month 0-Peru | 114 | 87 | 115 | 113 | 86 | 71 | 108 | 100 | 108 | 98 | 102
  CD4+-E M-N at Month 0-Total: number analyzed (Participants) | 336 | 243 | 337 | 264 | 202 | 184 | 322 | 313 | 318 | 275 | 290
  CD4+-E M-N at Month 0-Total | 200 | 144 | 197 | 161 | 123 | 103 | 182 | 170 | 187 | 154 | 170
  CD4+-E M-N at Month 0-USA: number analyzed (Participants) | 169 | 120 | 163 | 99 | 80 | 71 | 156 | 157 | 158 | 125 | 137
  CD4+-E M-N at Month 0-USA | 86 | 57 | 82 | 48 | 37 | 32 | 74 | 70 | 79 | 56 | 68
  CD4+-E M-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 61 | 8 | 18 | 14 | 24 | 21
  CD4+-E M-Y at Month 0-Peru | 1 | 28 | 0 | 2 | 29 | 44 | 7 | 15 | 7 | 17 | 13
  CD4+-E M-Y at Month 0-Total: number analyzed (Participants) | 22 | 115 | 21 | 94 | 156 | 174 | 36 | 45 | 40 | 83 | 68
  CD4+-E M-Y at Month 0-Total | 3 | 59 | 6 | 42 | 80 | 100 | 21 | 33 | 16 | 49 | 33
  CD4+-E M-Y at Month 0-USA: number analyzed (Participants) | 15 | 64 | 21 | 85 | 104 | 113 | 28 | 27 | 26 | 59 | 47
  CD4+-E M-Y at Month 0-USA | 2 | 31 | 6 | 40 | 51 | 56 | 14 | 18 | 9 | 32 | 20
  CD4+-N-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD4+-N-N at Month 0-Peru | 113 | 85 | 116 | 113 | 84 | 74 | 110 | 103 | 108 | 99 | 103
  CD4+-N-N at Month 0-Total: number analyzed (Participants) | 340 | 245 | 343 | 269 | 204 | 185 | 327 | 318 | 322 | 280 | 293
  CD4+-N-N at Month 0-Total | 214 | 152 | 214 | 169 | 127 | 111 | 196 | 192 | 201 | 168 | 181
  CD4+-N-N at Month 0-USA: number analyzed (Participants) | 171 | 121 | 167 | 102 | 81 | 72 | 160 | 160 | 161 | 128 | 139
  CD4+-N-N at Month 0-USA | 101 | 67 | 98 | 56 | 43 | 37 | 86 | 89 | 93 | 69 | 78
  CD4+-N-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD4+-N-Y at Month 0-Peru | 3 | 31 | 0 | 3 | 32 | 42 | 6 | 13 | 8 | 17 | 13
  CD4+-N-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 95 | 160 | 179 | 37 | 46 | 42 | 84 | 71
  CD4+-N-Y at Month 0-Total | 7 | 69 | 7 | 52 | 94 | 110 | 25 | 29 | 20 | 53 | 40
  CD4+-N-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 86 | 107 | 116 | 28 | 28 | 27 | 60 | 49
  CD4+-N-Y at Month 0-USA | 4 | 38 | 7 | 49 | 62 | 68 | 19 | 16 | 12 | 36 | 27
  CD4+-ORF3a6-N at Month 0-Peru: number analyzed (Participants) | 165 | 121 | 172 | 163 | 120 | 113 | 163 | 155 | 160 | 149 | 153
  CD4+-ORF3a6-N at Month 0-Peru | 65 | 49 | 65 | 63 | 48 | 40 | 61 | 58 | 63 | 52 | 59
  CD4+-ORF3a6-N at Month 0-Total: number analyzed (Participants) | 334 | 241 | 336 | 263 | 200 | 185 | 320 | 313 | 319 | 275 | 291
  CD4+-ORF3a6-N at Month 0-Total | 124 | 87 | 120 | 93 | 71 | 62 | 113 | 107 | 115 | 90 | 103
  CD4+-ORF3a6-N at Month 0-USA: number analyzed (Participants) | 169 | 120 | 164 | 100 | 80 | 72 | 157 | 158 | 159 | 126 | 138
  CD4+-ORF3a6-N at Month 0-USA | 59 | 38 | 55 | 30 | 23 | 22 | 52 | 49 | 52 | 38 | 44
  CD4+-ORF3a6-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 59 | 9 | 17 | 12 | 23 | 19
  CD4+-ORF3a6-Y at Month 0-Peru | 0 | 16 | 0 | 2 | 17 | 25 | 4 | 7 | 2 | 13 | 6
  CD4+-ORF3a6-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 94 | 157 | 172 | 37 | 44 | 38 | 82 | 66
  CD4+-ORF3a6-Y at Month 0-Total | 2 | 39 | 6 | 33 | 55 | 64 | 13 | 19 | 11 | 36 | 23
  CD4+-ORF3a6-Y at Month 0-USA: number analyzed (Participants) | 16 | 65 | 21 | 85 | 105 | 113 | 28 | 27 | 26 | 59 | 47
  CD4+-ORF3a6-Y at Month 0-USA | 2 | 23 | 6 | 31 | 38 | 39 | 9 | 12 | 9 | 23 | 17
  CD4+-ORF7a7b8-N at Month 0-Peru: number analyzed (Participants) | 167 | 124 | 174 | 165 | 123 | 112 | 165 | 156 | 160 | 150 | 153
  CD4+-ORF7a7b8-N at Month 0-Peru | 84 | 62 | 86 | 85 | 61 | 51 | 81 | 74 | 83 | 71 | 77
  CD4+-ORF7a7b8-N at Month 0-Total: number analyzed (Participants) | 333 | 242 | 336 | 263 | 202 | 183 | 320 | 311 | 318 | 274 | 290
  CD4+-ORF7a7b8-N at Month 0-Total | 138 | 92 | 138 | 111 | 79 | 70 | 127 | 118 | 133 | 107 | 120
  CD4+-ORF7a7b8-N at Month 0-USA: number analyzed (Participants) | 166 | 118 | 162 | 98 | 79 | 71 | 155 | 155 | 158 | 124 | 137
  CD4+-ORF7a7b8-N at Month 0-USA | 54 | 30 | 52 | 26 | 18 | 19 | 46 | 44 | 50 | 36 | 43
  CD4+-ORF7a7b8-Y at Month 0-Peru: number analyzed (Participants) | 7 | 50 | 0 | 9 | 51 | 62 | 9 | 18 | 14 | 24 | 21
  CD4+-ORF7a7b8-Y at Month 0-Peru | 2 | 24 | 0 | 1 | 25 | 35 | 5 | 12 | 3 | 15 | 9
  CD4+-ORF7a7b8-Y at Month 0-Total: number analyzed (Participants) | 23 | 114 | 20 | 93 | 154 | 173 | 36 | 45 | 38 | 82 | 66
  CD4+-ORF7a7b8-Y at Month 0-Total | 4 | 50 | 4 | 31 | 63 | 72 | 15 | 24 | 9 | 35 | 22
  CD4+-ORF7a7b8-Y at Month 0-USA: number analyzed (Participants) | 16 | 64 | 20 | 84 | 103 | 111 | 27 | 27 | 24 | 58 | 45
  CD4+-ORF7a7b8-Y at Month 0-USA | 2 | 26 | 4 | 30 | 38 | 37 | 10 | 12 | 6 | 20 | 13
  CD4+-S1-N at Month 0-Peru: number analyzed (Participants) | 166 | 121 | 173 | 164 | 120 | 112 | 164 | 155 | 159 | 150 | 152
  CD4+-S1-N at Month 0-Peru | 123 | 93 | 126 | 124 | 92 | 81 | 119 | 114 | 117 | 108 | 110
  CD4+-S1-N at Month 0-Total: number analyzed (Participants) | 337 | 242 | 340 | 265 | 200 | 183 | 324 | 315 | 319 | 278 | 290
  CD4+-S1-N at Month 0-Total | 225 | 162 | 222 | 181 | 136 | 119 | 208 | 203 | 207 | 178 | 185
  CD4+-S1-N at Month 0-USA: number analyzed (Participants) | 171 | 121 | 167 | 101 | 80 | 71 | 160 | 160 | 160 | 128 | 138
  CD4+-S1-N at Month 0-USA | 102 | 69 | 96 | 57 | 44 | 38 | 89 | 89 | 90 | 70 | 75
  CD4+-S1-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 61 | 9 | 18 | 14 | 23 | 21
  CD4+-S1-Y at Month 0-Peru | 3 | 33 | 0 | 2 | 34 | 45 | 7 | 12 | 9 | 18 | 16
  CD4+-S1-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 96 | 161 | 178 | 37 | 46 | 42 | 83 | 71
  CD4+-S1-Y at Month 0-Total | 6 | 69 | 9 | 50 | 95 | 112 | 23 | 28 | 24 | 53 | 46
  CD4+-S1-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 87 | 108 | 117 | 28 | 28 | 28 | 60 | 50
  CD4+-S1-Y at Month 0-USA | 3 | 36 | 9 | 48 | 61 | 67 | 16 | 16 | 15 | 35 | 30
  CD4+-S2-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD4+-S2-N at Month 0-Peru | 113 | 82 | 116 | 111 | 81 | 75 | 110 | 102 | 111 | 99 | 105
  CD4+-S2-N at Month 0-Total: number analyzed (Participants) | 341 | 246 | 344 | 269 | 204 | 185 | 328 | 319 | 322 | 281 | 293
  CD4+-S2-N at Month 0-Total | 213 | 150 | 211 | 165 | 124 | 112 | 199 | 186 | 200 | 167 | 179
  CD4+-S2-N at Month 0-USA: number analyzed (Participants) | 172 | 122 | 168 | 102 | 81 | 72 | 161 | 161 | 161 | 129 | 139
  CD4+-S2-N at Month 0-USA | 100 | 68 | 95 | 54 | 43 | 37 | 89 | 84 | 89 | 68 | 74
  CD4+-S2-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD4+-S2-Y at Month 0-Peru | 3 | 34 | 0 | 5 | 35 | 41 | 6 | 14 | 5 | 17 | 11
  CD4+-S2-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 96 | 161 | 180 | 37 | 46 | 43 | 84 | 72
  CD4+-S2-Y at Month 0-Total | 6 | 69 | 8 | 54 | 95 | 107 | 20 | 33 | 19 | 52 | 40
  CD4+-S2-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 87 | 108 | 117 | 28 | 28 | 28 | 60 | 50
  CD4+-S2-Y at Month 0-USA | 3 | 35 | 8 | 49 | 60 | 66 | 14 | 19 | 14 | 35 | 29
  CD4+-Spike-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD4+-Spike-N at Month 0-Peru | 131 | 98 | 135 | 130 | 97 | 88 | 128 | 121 | 126 | 117 | 119
  CD4+-Spike-N at Month 0-Total: number analyzed (Participants) | 341 | 246 | 344 | 269 | 204 | 185 | 328 | 319 | 322 | 281 | 293
  CD4+-Spike-N at Month 0-Total | 244 | 174 | 242 | 193 | 146 | 131 | 227 | 219 | 226 | 196 | 203
  CD4+-Spike-N at Month 0-USA: number analyzed (Participants) | 172 | 122 | 168 | 102 | 81 | 72 | 161 | 161 | 161 | 129 | 139
  CD4+-Spike-N at Month 0-USA | 113 | 76 | 107 | 63 | 49 | 43 | 99 | 98 | 100 | 79 | 84
  CD4+-Spike-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD4+-Spike-Y at Month 0-Peru | 4 | 37 | 0 | 5 | 38 | 47 | 7 | 14 | 9 | 18 | 16
  CD4+-Spike-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 96 | 161 | 180 | 37 | 46 | 43 | 84 | 72
  CD4+-Spike-Y at Month 0-Total | 8 | 78 | 10 | 59 | 106 | 121 | 25 | 33 | 26 | 56 | 49
  CD4+-Spike-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 87 | 108 | 117 | 28 | 28 | 28 | 60 | 50
  CD4+-Spike-Y at Month 0-USA | 4 | 41 | 10 | 54 | 68 | 74 | 18 | 19 | 17 | 38 | 33
  CD8+-Any COV2-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD8+-Any COV2-N at Month 0-Peru | 117 | 88 | 122 | 117 | 87 | 89 | 118 | 111 | 115 | 109 | 111
  CD8+-Any COV2-N at Month 0-Total: number analyzed (Participants) | 340 | 245 | 343 | 269 | 204 | 184 | 327 | 318 | 321 | 280 | 292
  CD8+-Any COV2-N at Month 0-Total | 218 | 165 | 221 | 176 | 138 | 131 | 211 | 203 | 210 | 191 | 193
  CD8+-Any COV2-N at Month 0-USA: number analyzed (Participants) | 171 | 121 | 167 | 102 | 81 | 71 | 160 | 160 | 160 | 128 | 138
  CD8+-Any COV2-N at Month 0-USA | 101 | 77 | 99 | 59 | 51 | 42 | 93 | 92 | 95 | 82 | 82
  CD8+-Any COV2-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD8+-Any COV2-Y at Month 0-Peru | 5 | 34 | 0 | 5 | 35 | 33 | 4 | 11 | 7 | 13 | 11
  CD8+-Any COV2-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 95 | 160 | 180 | 37 | 46 | 43 | 84 | 72
  CD8+-Any COV2-Y at Month 0-Total | 14 | 67 | 11 | 56 | 94 | 101 | 21 | 29 | 22 | 41 | 39
  CD8+-Any COV2-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 86 | 107 | 117 | 28 | 28 | 28 | 60 | 50
  CD8+-Any COV2-Y at Month 0-USA | 9 | 33 | 11 | 51 | 59 | 68 | 17 | 18 | 15 | 28 | 28
  CD8+-E M-N at Month 0-Peru: number analyzed (Participants) | 168 | 124 | 175 | 166 | 123 | 113 | 166 | 157 | 161 | 151 | 154
  CD8+-E M-N at Month 0-Peru | 13 | 11 | 13 | 13 | 11 | 9 | 12 | 12 | 12 | 11 | 12
  CD8+-E M-N at Month 0-Total: number analyzed (Participants) | 335 | 242 | 337 | 266 | 203 | 184 | 321 | 313 | 318 | 275 | 291
  CD8+-E M-N at Month 0-Total | 29 | 24 | 28 | 24 | 20 | 17 | 26 | 28 | 26 | 21 | 24
  CD8+-E M-N at Month 0-USA: number analyzed (Participants) | 167 | 118 | 162 | 100 | 80 | 71 | 155 | 156 | 157 | 124 | 137
  CD8+-E M-N at Month 0-USA | 16 | 13 | 15 | 11 | 9 | 8 | 14 | 16 | 14 | 10 | 12
  CD8+-E M-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 62 | 9 | 18 | 14 | 24 | 21
  CD8+-E M-Y at Month 0-Peru | 0 | 2 | 0 | 0 | 2 | 4 | 1 | 1 | 1 | 2 | 1
  CD8+-E M-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 92 | 155 | 174 | 37 | 45 | 40 | 83 | 67
  CD8+-E M-Y at Month 0-Total | 1 | 6 | 2 | 6 | 10 | 13 | 4 | 2 | 4 | 9 | 6
  CD8+-E M-Y at Month 0-USA: number analyzed (Participants) | 16 | 65 | 21 | 83 | 103 | 112 | 28 | 27 | 26 | 59 | 46
  CD8+-E M-Y at Month 0-USA | 1 | 4 | 2 | 6 | 8 | 9 | 3 | 1 | 3 | 7 | 5
  CD8+-N-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD8+-N-N at Month 0-Peru | 103 | 76 | 108 | 103 | 75 | 75 | 104 | 97 | 101 | 95 | 97
  CD8+-N-N at Month 0-Total: number analyzed (Participants) | 339 | 244 | 342 | 269 | 204 | 184 | 326 | 317 | 321 | 279 | 292
  CD8+-N-N at Month 0-Total | 188 | 143 | 191 | 152 | 117 | 111 | 182 | 174 | 183 | 164 | 168
  CD8+-N-N at Month 0-USA: number analyzed (Participants) | 170 | 120 | 166 | 102 | 81 | 71 | 159 | 159 | 160 | 127 | 138
  CD8+-N-N at Month 0-USA | 85 | 67 | 83 | 49 | 42 | 36 | 78 | 77 | 82 | 69 | 71
  CD8+-N-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD8+-N-Y at Month 0-Peru | 5 | 32 | 0 | 5 | 33 | 33 | 4 | 11 | 7 | 13 | 11
  CD8+-N-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 94 | 159 | 179 | 37 | 46 | 42 | 84 | 71
  CD8+-N-Y at Month 0-Total | 12 | 57 | 9 | 48 | 83 | 89 | 18 | 26 | 17 | 36 | 32
  CD8+-N-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 85 | 106 | 116 | 28 | 28 | 27 | 60 | 49
  CD8+-N-Y at Month 0-USA | 7 | 25 | 9 | 43 | 50 | 56 | 14 | 15 | 10 | 23 | 21
  CD8+-ORF3a6-N at Month 0-Peru: number analyzed (Participants) | 167 | 123 | 174 | 165 | 122 | 113 | 165 | 157 | 160 | 151 | 153
  CD8+-ORF3a6-N at Month 0-Peru | 46 | 34 | 50 | 47 | 33 | 33 | 48 | 44 | 45 | 46 | 44
  CD8+-ORF3a6-N at Month 0-Total: number analyzed (Participants) | 335 | 242 | 337 | 265 | 202 | 184 | 321 | 314 | 318 | 276 | 290
  CD8+-ORF3a6-N at Month 0-Total | 73 | 52 | 77 | 61 | 44 | 43 | 75 | 68 | 69 | 66 | 66
  CD8+-ORF3a6-N at Month 0-USA: number analyzed (Participants) | 168 | 119 | 163 | 100 | 80 | 71 | 156 | 157 | 158 | 125 | 137
  CD8+-ORF3a6-N at Month 0-USA | 27 | 18 | 27 | 14 | 11 | 10 | 27 | 24 | 24 | 20 | 22
  CD8+-ORF3a6-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 61 | 9 | 17 | 14 | 23 | 21
  CD8+-ORF3a6-Y at Month 0-Peru | 4 | 16 | 0 | 3 | 17 | 17 | 2 | 6 | 5 | 4 | 6
  CD8+-ORF3a6-Y at Month 0-Total: number analyzed (Participants) | 23 | 116 | 21 | 93 | 156 | 174 | 37 | 44 | 40 | 82 | 68
  CD8+-ORF3a6-Y at Month 0-Total | 7 | 28 | 3 | 19 | 36 | 37 | 5 | 12 | 11 | 14 | 14
  CD8+-ORF3a6-Y at Month 0-USA: number analyzed (Participants) | 16 | 65 | 21 | 84 | 104 | 113 | 28 | 27 | 26 | 59 | 47
  CD8+-ORF3a6-Y at Month 0-USA | 3 | 12 | 3 | 16 | 19 | 20 | 3 | 6 | 6 | 10 | 8
  CD8+-ORF7a7b8-N at Month 0-Peru: number analyzed (Participants) | 167 | 124 | 174 | 165 | 123 | 112 | 165 | 156 | 160 | 150 | 153
  CD8+-ORF7a7b8-N at Month 0-Peru | 49 | 35 | 51 | 48 | 34 | 34 | 49 | 44 | 46 | 47 | 46
  CD8+-ORF7a7b8-N at Month 0-Total: number analyzed (Participants) | 331 | 240 | 334 | 262 | 201 | 181 | 318 | 309 | 316 | 272 | 288
  CD8+-ORF7a7b8-N at Month 0-Total | 67 | 49 | 71 | 59 | 44 | 38 | 66 | 60 | 59 | 60 | 57
  CD8+-ORF7a7b8-N at Month 0-USA: number analyzed (Participants) | 164 | 116 | 160 | 97 | 78 | 69 | 153 | 153 | 156 | 122 | 135
  CD8+-ORF7a7b8-N at Month 0-USA | 18 | 14 | 20 | 11 | 10 | 4 | 17 | 16 | 13 | 13 | 11
  CD8+-ORF7a7b8-Y at Month 0-Peru: number analyzed (Participants) | 7 | 50 | 0 | 9 | 51 | 62 | 9 | 18 | 14 | 24 | 21
  CD8+-ORF7a7b8-Y at Month 0-Peru | 2 | 16 | 0 | 3 | 17 | 17 | 2 | 7 | 5 | 4 | 5
  CD8+-ORF7a7b8-Y at Month 0-Total: number analyzed (Participants) | 23 | 114 | 20 | 92 | 153 | 173 | 36 | 45 | 38 | 82 | 66
  CD8+-ORF7a7b8-Y at Month 0-Total | 4 | 22 | 0 | 12 | 27 | 33 | 5 | 11 | 12 | 11 | 14
  CD8+-ORF7a7b8-Y at Month 0-USA: number analyzed (Participants) | 16 | 64 | 20 | 83 | 102 | 111 | 27 | 27 | 24 | 58 | 45
  CD8+-ORF7a7b8-Y at Month 0-USA | 2 | 6 | 0 | 9 | 10 | 16 | 3 | 4 | 7 | 7 | 9
  CD8+-S1-N at Month 0-Peru: number analyzed (Participants) | 167 | 122 | 174 | 165 | 121 | 112 | 165 | 156 | 159 | 151 | 152
  CD8+-S1-N at Month 0-Peru | 42 | 33 | 42 | 42 | 33 | 31 | 40 | 39 | 39 | 38 | 38
  CD8+-S1-N at Month 0-Total: number analyzed (Participants) | 337 | 242 | 340 | 266 | 201 | 182 | 324 | 315 | 318 | 278 | 289
  CD8+-S1-N at Month 0-Total | 71 | 52 | 69 | 52 | 42 | 42 | 63 | 63 | 65 | 63 | 59
  CD8+-S1-N at Month 0-USA: number analyzed (Participants) | 170 | 120 | 166 | 101 | 80 | 70 | 159 | 159 | 159 | 127 | 137
  CD8+-S1-N at Month 0-USA | 29 | 19 | 27 | 10 | 9 | 11 | 23 | 24 | 26 | 25 | 21
  CD8+-S1-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 62 | 9 | 18 | 15 | 23 | 22
  CD8+-S1-Y at Month 0-Peru | 0 | 9 | 0 | 0 | 9 | 11 | 2 | 3 | 3 | 4 | 4
  CD8+-S1-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 95 | 160 | 179 | 37 | 46 | 43 | 83 | 72
  CD8+-S1-Y at Month 0-Total | 0 | 19 | 2 | 19 | 29 | 29 | 8 | 8 | 6 | 8 | 12
  CD8+-S1-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 86 | 107 | 117 | 28 | 28 | 28 | 60 | 50
  CD8+-S1-Y at Month 0-USA | 0 | 10 | 2 | 19 | 20 | 18 | 6 | 5 | 3 | 4 | 8
  CD8+-S2-N at Month 0-Peru: number analyzed (Participants) | 168 | 124 | 175 | 166 | 123 | 113 | 166 | 158 | 160 | 151 | 153
  CD8+-S2-N at Month 0-Peru | 18 | 14 | 18 | 18 | 14 | 15 | 18 | 18 | 18 | 15 | 18
  CD8+-S2-N at Month 0-Total: number analyzed (Participants) | 339 | 245 | 342 | 268 | 204 | 184 | 326 | 318 | 320 | 279 | 291
  CD8+-S2-N at Month 0-Total | 30 | 24 | 30 | 27 | 23 | 23 | 28 | 29 | 30 | 26 | 28
  CD8+-S2-N at Month 0-USA: number analyzed (Participants) | 171 | 121 | 167 | 102 | 81 | 71 | 160 | 160 | 160 | 128 | 138
  CD8+-S2-N at Month 0-USA | 12 | 10 | 12 | 9 | 9 | 8 | 10 | 11 | 12 | 11 | 10
  CD8+-S2-Y at Month 0-Peru: number analyzed (Participants) | 7 | 51 | 0 | 9 | 52 | 62 | 9 | 17 | 15 | 24 | 22
  CD8+-S2-Y at Month 0-Peru | 0 | 4 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 3 | 0
  CD8+-S2-Y at Month 0-Total: number analyzed (Participants) | 24 | 118 | 21 | 95 | 159 | 179 | 37 | 45 | 43 | 84 | 72
  CD8+-S2-Y at Month 0-Total | 0 | 6 | 0 | 3 | 7 | 7 | 2 | 1 | 0 | 4 | 2
  CD8+-S2-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 86 | 107 | 117 | 28 | 28 | 28 | 60 | 50
  CD8+-S2-Y at Month 0-USA | 0 | 2 | 0 | 3 | 3 | 4 | 2 | 1 | 0 | 1 | 2
  CD8+-Spike-N at Month 0-Peru: number analyzed (Participants) | 169 | 124 | 176 | 167 | 123 | 113 | 167 | 158 | 161 | 152 | 154
  CD8+-Spike-N at Month 0-Peru | 47 | 37 | 47 | 47 | 37 | 35 | 45 | 44 | 44 | 42 | 43
  CD8+-Spike-N at Month 0-Total: number analyzed (Participants) | 340 | 245 | 343 | 269 | 204 | 184 | 327 | 318 | 321 | 280 | 292
  CD8+-Spike-N at Month 0-Total | 82 | 61 | 80 | 62 | 51 | 50 | 73 | 73 | 76 | 72 | 70
  CD8+-Spike-N at Month 0-USA: number analyzed (Participants) | 171 | 121 | 167 | 102 | 81 | 71 | 160 | 160 | 160 | 128 | 138
  CD8+-Spike-N at Month 0-USA | 35 | 24 | 33 | 15 | 14 | 15 | 28 | 29 | 32 | 30 | 27
  CD8+-Spike-Y at Month 0-Peru: number analyzed (Participants) | 7 | 52 | 0 | 9 | 53 | 63 | 9 | 18 | 15 | 24 | 22
  CD8+-Spike-Y at Month 0-Peru | 0 | 10 | 0 | 0 | 10 | 12 | 2 | 3 | 3 | 5 | 4
  CD8+-Spike-Y at Month 0-Total: number analyzed (Participants) | 24 | 119 | 21 | 95 | 160 | 180 | 37 | 46 | 43 | 84 | 72
  CD8+-Spike-Y at Month 0-Total | 0 | 21 | 2 | 20 | 31 | 32 | 9 | 9 | 6 | 10 | 12
  CD8+-Spike-Y at Month 0-USA: number analyzed (Participants) | 17 | 67 | 21 | 86 | 107 | 117 | 28 | 28 | 28 | 60 | 50
  CD8+-Spike-Y at Month 0-USA | 0 | 11 | 2 | 20 | 21 | 20 | 7 | 6 | 3 | 5 | 8

59. Primary Outcome: SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude (ICS) by Region and Comorbidity Group Among America Cohort
Description: Flow cytometry was used to examine SARS-CoV-2 specific CD4+ and CD8+ T-cell responses using an intracellular cytokine staining (ICS). Positive calls will be made using Fisher's exact positivity test for all the markers. The magnitudes are % T cells expressing IFN-g/IL-2.
  The table summarized SARS-CoV-2-specific CD4+ and CD8+ T Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and Comorbidity Group among America Cohort
Time Frame: Measured at Months 0
Population: American Population with positive responders (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: % T cells expressing IFN-g/IL-2
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
% T cells expressing IFN-g/IL-2
  CD4+-Any COV2-N at Month 0-Peru: number analyzed (Participants) | 139 | 105 | 143 | 138 | 104 | 91 | 135 | 128 | 132 | 124 | 125
  CD4+-Any COV2-N at Month 0-Peru | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.2] | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.2] | 0.6 [0.4 to 1.3] | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.3] | 0.7 [0.4 to 1.3] | 0.6 [0.4 to 1.3] | 0.7 [0.4 to 1.3]
  CD4+-Any COV2-N at Month 0-Total: number analyzed (Participants) | 263 | 189 | 261 | 209 | 160 | 138 | 245 | 236 | 242 | 212 | 217
  CD4+-Any COV2-N at Month 0-Total | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.2] | 0.6 [0.3 to 1.1] | 0.5 [0.3 to 1.2] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.2]
  CD4+-Any COV2-N at Month 0-USA: number analyzed (Participants) | 124 | 84 | 118 | 71 | 56 | 47 | 110 | 108 | 110 | 88 | 92
  CD4+-Any COV2-N at Month 0-USA | 0.5 [0.3 to 1] | 0.5 [0.3 to 0.9] | 0.5 [0.3 to 1] | 0.5 [0.3 to 0.9] | 0.5 [0.3 to 0.8] | 0.4 [0.2 to 0.9] | 0.5 [0.3 to 0.9] | 0.5 [0.3 to 1] | 0.5 [0.3 to 1] | 0.4 [0.3 to 0.9] | 0.5 [0.3 to 1]
  CD4+-Any COV2-Y at Month 0-Peru: number analyzed (Participants) | 4 | 38 | 0 | 5 | 39 | 52 | 8 | 15 | 11 | 19 | 18
  CD4+-Any COV2-Y at Month 0-Peru | 0.3 [0.3 to 0.4] | 0.9 [0.4 to 1.4] |  | 0.2 [0.2 to 0.5] | 0.9 [0.4 to 1.4] | 0.9 [0.5 to 1.3] | 0.9 [0.5 to 1.2] | 1.1 [0.7 to 1.6] | 0.6 [0.3 to 1] | 0.9 [0.7 to 1.3] | 0.6 [0.3 to 1.2]
  CD4+-Any COV2-Y at Month 0-Total: number analyzed (Participants) | 9 | 83 | 11 | 63 | 112 | 134 | 27 | 36 | 30 | 60 | 55
  CD4+-Any COV2-Y at Month 0-Total | 0.3 [0.3 to 0.9] | 0.7 [0.3 to 1.3] | 0.4 [0.3 to 1.2] | 0.6 [0.3 to 1.1] | 0.7 [0.3 to 1.2] | 0.7 [0.4 to 1.1] | 0.9 [0.3 to 1.1] | 0.8 [0.5 to 1.2] | 0.6 [0.3 to 1.1] | 0.9 [0.5 to 1.2] | 0.6 [0.3 to 1]
  CD4+-Any COV2-Y at Month 0-USA: number analyzed (Participants) | 5 | 45 | 11 | 58 | 73 | 82 | 19 | 21 | 19 | 41 | 37
  CD4+-Any COV2-Y at Month 0-USA | 0.5 [0.3 to 1.1] | 0.7 [0.3 to 1.2] | 0.4 [0.3 to 1.2] | 0.6 [0.3 to 1.1] | 0.6 [0.3 to 1.1] | 0.6 [0.4 to 1] | 1 [0.3 to 1.1] | 0.8 [0.5 to 1.1] | 0.6 [0.3 to 1.1] | 0.8 [0.5 to 1.1] | 0.6 [0.3 to 1]
  CD4+-E M-N at Month 0-Peru: number analyzed (Participants) | 114 | 87 | 115 | 113 | 86 | 71 | 108 | 100 | 108 | 98 | 102
  CD4+-E M-N at Month 0-Peru | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M-N at Month 0-Total: number analyzed (Participants) | 200 | 144 | 197 | 161 | 123 | 103 | 182 | 170 | 187 | 154 | 170
  CD4+-E M-N at Month 0-Total | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M-N at Month 0-USA: number analyzed (Participants) | 86 | 57 | 82 | 48 | 37 | 32 | 74 | 70 | 79 | 56 | 68
  CD4+-E M-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-E M-Y at Month 0-Peru: number analyzed (Participants) | 1 | 28 | 0 | 2 | 29 | 44 | 7 | 15 | 7 | 17 | 13
  CD4+-E M-Y at Month 0-Peru | 0.3 [0.3 to 0.3] | 0.3 [0.1 to 0.4] |  | 0.2 [0.2 to 0.3] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.4]
  CD4+-E M-Y at Month 0-Total: number analyzed (Participants) | 3 | 59 | 6 | 42 | 80 | 100 | 21 | 33 | 16 | 49 | 33
  CD4+-E M-Y at Month 0-Total | 0.3 [0.2 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-E M-Y at Month 0-USA: number analyzed (Participants) | 2 | 31 | 6 | 40 | 51 | 56 | 14 | 18 | 9 | 32 | 20
  CD4+-E M-Y at Month 0-USA | 0.2 [0.2 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.2 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD4+-N-N at Month 0-Peru: number analyzed (Participants) | 113 | 85 | 116 | 113 | 84 | 74 | 110 | 103 | 108 | 99 | 103
  CD4+-N-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N-N at Month 0-Total: number analyzed (Participants) | 214 | 152 | 214 | 169 | 127 | 111 | 196 | 192 | 201 | 168 | 181
  CD4+-N-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N-N at Month 0-USA: number analyzed (Participants) | 101 | 67 | 98 | 56 | 43 | 37 | 86 | 89 | 93 | 69 | 78
  CD4+-N-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD4+-N-Y at Month 0-Peru: number analyzed (Participants) | 3 | 31 | 0 | 3 | 32 | 42 | 6 | 13 | 8 | 17 | 13
  CD4+-N-Y at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] |  | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N-Y at Month 0-Total: number analyzed (Participants) | 7 | 69 | 7 | 52 | 94 | 110 | 25 | 29 | 20 | 53 | 40
  CD4+-N-Y at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-N-Y at Month 0-USA: number analyzed (Participants) | 4 | 38 | 7 | 49 | 62 | 68 | 19 | 16 | 12 | 36 | 27
  CD4+-N-Y at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  CD4+-ORF3a6-N at Month 0-Peru: number analyzed (Participants) | 65 | 49 | 65 | 63 | 48 | 40 | 61 | 58 | 63 | 52 | 59
  CD4+-ORF3a6-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6-N at Month 0-Total: number analyzed (Participants) | 124 | 87 | 120 | 93 | 71 | 62 | 113 | 107 | 115 | 90 | 103
  CD4+-ORF3a6-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6-N at Month 0-USA: number analyzed (Participants) | 59 | 38 | 55 | 30 | 23 | 22 | 52 | 49 | 52 | 38 | 44
  CD4+-ORF3a6-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF3a6-Y at Month 0-Peru: number analyzed (Participants) | 0 | 16 | 0 | 2 | 17 | 25 | 4 | 7 | 2 | 13 | 6
  CD4+-ORF3a6-Y at Month 0-Peru |  | 0.1 [0.1 to 0.2] |  | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD4+-ORF3a6-Y at Month 0-Total: number analyzed (Participants) | 2 | 39 | 6 | 33 | 55 | 64 | 13 | 19 | 11 | 36 | 23
  CD4+-ORF3a6-Y at Month 0-Total | 0.6 [0.4 to 0.8] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3]
  CD4+-ORF3a6-Y at Month 0-USA: number analyzed (Participants) | 2 | 23 | 6 | 31 | 38 | 39 | 9 | 12 | 9 | 23 | 17
  CD4+-ORF3a6-Y at Month 0-USA | 0.6 [0.4 to 0.8] | 0.1 [0.1 to 0.2] | 0.2 [0.2 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8-N at Month 0-Peru: number analyzed (Participants) | 84 | 62 | 86 | 85 | 61 | 51 | 81 | 74 | 83 | 71 | 77
  CD4+-ORF7a7b8-N at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8-N at Month 0-Total: number analyzed (Participants) | 138 | 92 | 138 | 111 | 79 | 70 | 127 | 118 | 133 | 107 | 120
  CD4+-ORF7a7b8-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8-N at Month 0-USA: number analyzed (Participants) | 54 | 30 | 52 | 26 | 18 | 19 | 46 | 44 | 50 | 36 | 43
  CD4+-ORF7a7b8-N at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-ORF7a7b8-Y at Month 0-Peru: number analyzed (Participants) | 2 | 24 | 0 | 1 | 25 | 35 | 5 | 12 | 3 | 15 | 9
  CD4+-ORF7a7b8-Y at Month 0-Peru | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2] |  | 0 [0 to 0] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.2]
  CD4+-ORF7a7b8-Y at Month 0-Total: number analyzed (Participants) | 4 | 50 | 4 | 31 | 63 | 72 | 15 | 24 | 9 | 35 | 22
  CD4+-ORF7a7b8-Y at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1]
  CD4+-ORF7a7b8-Y at Month 0-USA: number analyzed (Participants) | 2 | 26 | 4 | 30 | 38 | 37 | 10 | 12 | 6 | 20 | 13
  CD4+-ORF7a7b8-Y at Month 0-USA | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  CD4+-S1-N at Month 0-Peru: number analyzed (Participants) | 123 | 93 | 126 | 124 | 92 | 81 | 119 | 114 | 117 | 108 | 110
  CD4+-S1-N at Month 0-Peru | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  CD4+-S1-N at Month 0-Total: number analyzed (Participants) | 225 | 162 | 222 | 181 | 136 | 119 | 208 | 203 | 207 | 178 | 185
  CD4+-S1-N at Month 0-Total | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4]
  CD4+-S1-N at Month 0-USA: number analyzed (Participants) | 102 | 69 | 96 | 57 | 44 | 38 | 89 | 89 | 90 | 70 | 75
  CD4+-S1-N at Month 0-USA | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD4+-S1-Y at Month 0-Peru: number analyzed (Participants) | 3 | 33 | 0 | 2 | 34 | 45 | 7 | 12 | 9 | 18 | 16
  CD4+-S1-Y at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.4] |  | 0.4 [0.2 to 0.5] | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0.2 [0.2 to 0.3] | 0.4 [0.3 to 0.5] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.4]
  CD4+-S1-Y at Month 0-Total: number analyzed (Participants) | 6 | 69 | 9 | 50 | 95 | 112 | 23 | 28 | 24 | 53 | 46
  CD4+-S1-Y at Month 0-Total | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3]
  CD4+-S1-Y at Month 0-USA: number analyzed (Participants) | 3 | 36 | 9 | 48 | 61 | 67 | 16 | 16 | 15 | 35 | 30
  CD4+-S1-Y at Month 0-USA | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD4+-S2-N at Month 0-Peru: number analyzed (Participants) | 113 | 82 | 116 | 111 | 81 | 75 | 110 | 102 | 111 | 99 | 105
  CD4+-S2-N at Month 0-Peru | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  CD4+-S2-N at Month 0-Total: number analyzed (Participants) | 213 | 150 | 211 | 165 | 124 | 112 | 199 | 186 | 200 | 167 | 179
  CD4+-S2-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2-N at Month 0-USA: number analyzed (Participants) | 100 | 68 | 95 | 54 | 43 | 37 | 89 | 84 | 89 | 68 | 74
  CD4+-S2-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2-Y at Month 0-Peru: number analyzed (Participants) | 3 | 34 | 0 | 5 | 35 | 41 | 6 | 14 | 5 | 17 | 11
  CD4+-S2-Y at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] |  | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2-Y at Month 0-Total: number analyzed (Participants) | 6 | 69 | 8 | 54 | 95 | 107 | 20 | 33 | 19 | 52 | 40
  CD4+-S2-Y at Month 0-Total | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD4+-S2-Y at Month 0-USA: number analyzed (Participants) | 3 | 35 | 8 | 49 | 60 | 66 | 14 | 19 | 14 | 35 | 29
  CD4+-S2-Y at Month 0-USA | 0 [0 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2]
  CD4+-Spike-N at Month 0-Peru: number analyzed (Participants) | 131 | 98 | 135 | 130 | 97 | 88 | 128 | 121 | 126 | 117 | 119
  CD4+-Spike-N at Month 0-Peru | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.6]
  CD4+-Spike-N at Month 0-Total: number analyzed (Participants) | 244 | 174 | 242 | 193 | 146 | 131 | 227 | 219 | 226 | 196 | 203
  CD4+-Spike-N at Month 0-Total | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.5]
  CD4+-Spike-N at Month 0-USA: number analyzed (Participants) | 113 | 76 | 107 | 63 | 49 | 43 | 99 | 98 | 100 | 79 | 84
  CD4+-Spike-N at Month 0-USA | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4]
  CD4+-Spike-Y at Month 0-Peru: number analyzed (Participants) | 4 | 37 | 0 | 5 | 38 | 47 | 7 | 14 | 9 | 18 | 16
  CD4+-Spike-Y at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.4 [0.2 to 0.7] |  | 0.1 [0.1 to 0.2] | 0.4 [0.2 to 0.7] | 0.4 [0.3 to 0.6] | 0.3 [0.3 to 0.5] | 0.5 [0.4 to 0.6] | 0.3 [0.2 to 0.6] | 0.5 [0.3 to 0.7] | 0.3 [0.2 to 0.6]
  CD4+-Spike-Y at Month 0-Total: number analyzed (Participants) | 8 | 78 | 10 | 59 | 106 | 121 | 25 | 33 | 26 | 56 | 49
  CD4+-Spike-Y at Month 0-Total | 0.1 [0.1 to 0.2] | 0.3 [0.2 to 0.6] | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.6] | 0.3 [0.1 to 0.5] | 0.4 [0.2 to 0.6] | 0.3 [0.2 to 0.5] | 0.4 [0.2 to 0.6] | 0.3 [0.2 to 0.5]
  CD4+-Spike-Y at Month 0-USA: number analyzed (Participants) | 4 | 41 | 10 | 54 | 68 | 74 | 18 | 19 | 17 | 38 | 33
  CD4+-Spike-Y at Month 0-USA | 0.2 [0.1 to 0.2] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.5] | 0.3 [0.1 to 0.5] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.5] | 0.3 [0.2 to 0.5] | 0.3 [0.1 to 0.4] | 0.3 [0.2 to 0.5] | 0.3 [0.1 to 0.5]
  CD8+-Any COV2-N at Month 0-Peru: number analyzed (Participants) | 117 | 88 | 122 | 117 | 87 | 89 | 118 | 111 | 115 | 109 | 111
  CD8+-Any COV2-N at Month 0-Peru | 0.5 [0.2 to 1.3] | 0.5 [0.2 to 1.3] | 0.5 [0.2 to 1.2] | 0.5 [0.2 to 1.3] | 0.5 [0.2 to 1.3] | 0.4 [0.2 to 0.9] | 0.5 [0.2 to 1.3] | 0.5 [0.2 to 1.1] | 0.5 [0.2 to 1.1] | 0.5 [0.2 to 1.1] | 0.5 [0.2 to 1.2]
  CD8+-Any COV2-N at Month 0-Total: number analyzed (Participants) | 218 | 165 | 221 | 176 | 138 | 131 | 211 | 203 | 210 | 191 | 193
  CD8+-Any COV2-N at Month 0-Total | 0.4 [0.2 to 0.9] | 0.3 [0.2 to 0.9] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 1.1] | 0.4 [0.2 to 1] | 0.4 [0.2 to 0.8] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 0.9] | 0.4 [0.2 to 0.9]
  CD8+-Any COV2-N at Month 0-USA: number analyzed (Participants) | 101 | 77 | 99 | 59 | 51 | 42 | 93 | 92 | 95 | 82 | 82
  CD8+-Any COV2-N at Month 0-USA | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.8] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.6] | 0.3 [0.2 to 0.7]
  CD8+-Any COV2-Y at Month 0-Peru: number analyzed (Participants) | 5 | 34 | 0 | 5 | 35 | 33 | 4 | 11 | 7 | 13 | 11
  CD8+-Any COV2-Y at Month 0-Peru | 0.4 [0.3 to 0.6] | 0.6 [0.4 to 1.1] |  | 0.4 [0.4 to 0.6] | 0.5 [0.4 to 1.1] | 0.9 [0.5 to 2.5] | 1 [0.9 to 1] | 1.1 [0.7 to 7.9] | 0.8 [0.6 to 1.6] | 0.6 [0.3 to 2.3] | 0.6 [0.4 to 1.1]
  CD8+-Any COV2-Y at Month 0-Total: number analyzed (Participants) | 14 | 67 | 11 | 56 | 94 | 101 | 21 | 29 | 22 | 41 | 39
  CD8+-Any COV2-Y at Month 0-Total | 0.2 [0.1 to 0.4] | 0.5 [0.2 to 0.9] | 0.2 [0.1 to 0.3] | 0.4 [0.1 to 0.7] | 0.4 [0.2 to 0.8] | 0.4 [0.2 to 1] | 0.4 [0.2 to 0.8] | 0.5 [0.2 to 1.1] | 0.5 [0.1 to 1.2] | 0.5 [0.2 to 1.1] | 0.3 [0.1 to 0.8]
  CD8+-Any COV2-Y at Month 0-USA: number analyzed (Participants) | 9 | 33 | 11 | 51 | 59 | 68 | 17 | 18 | 15 | 28 | 28
  CD8+-Any COV2-Y at Month 0-USA | 0.1 [0.1 to 0.2] | 0.4 [0.1 to 0.8] | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.7] | 0.3 [0.1 to 0.7] | 0.3 [0.1 to 0.7] | 0.3 [0.2 to 0.7] | 0.3 [0.2 to 0.7] | 0.2 [0.1 to 0.7] | 0.4 [0.1 to 0.8] | 0.3 [0.1 to 0.7]
  CD8+-E M-N at Month 0-Peru: number analyzed (Participants) | 13 | 11 | 13 | 13 | 11 | 9 | 12 | 12 | 12 | 11 | 12
  CD8+-E M-N at Month 0-Peru | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2]
  CD8+-E M-N at Month 0-Total: number analyzed (Participants) | 29 | 24 | 28 | 24 | 20 | 17 | 26 | 28 | 26 | 21 | 24
  CD8+-E M-N at Month 0-Total | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2]
  CD8+-E M-N at Month 0-USA: number analyzed (Participants) | 16 | 13 | 15 | 11 | 9 | 8 | 14 | 16 | 14 | 10 | 12
  CD8+-E M-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.5] | 0.1 [0.1 to 0.7] | 0.2 [0.1 to 0.7] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.6] | 0.1 [0.1 to 0.3]
  CD8+-E M-Y at Month 0-Peru: number analyzed (Participants) | 0 | 2 | 0 | 0 | 2 | 4 | 1 | 1 | 1 | 2 | 1
  CD8+-E M-Y at Month 0-Peru |  | 0.2 [0.2 to 0.3] |  |  | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2] | 0.3 [0.3 to 0.3] | 0.2 [0.2 to 0.2] | 0.3 [0.3 to 0.3]
  CD8+-E M-Y at Month 0-Total: number analyzed (Participants) | 1 | 6 | 2 | 6 | 10 | 13 | 4 | 2 | 4 | 9 | 6
  CD8+-E M-Y at Month 0-Total | 0 [0 to 0] | 0.1 [0 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-E M-Y at Month 0-USA: number analyzed (Participants) | 1 | 4 | 2 | 6 | 8 | 9 | 3 | 1 | 3 | 7 | 5
  CD8+-E M-Y at Month 0-USA | 0 [0 to 0] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0 to 0.2]
  CD8+-N-N at Month 0-Peru: number analyzed (Participants) | 103 | 76 | 108 | 103 | 75 | 75 | 104 | 97 | 101 | 95 | 97
  CD8+-N-N at Month 0-Peru | 0.3 [0.1 to 0.7] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.7]
  CD8+-N-N at Month 0-Total: number analyzed (Participants) | 188 | 143 | 191 | 152 | 117 | 111 | 182 | 174 | 183 | 164 | 168
  CD8+-N-N at Month 0-Total | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.5]
  CD8+-N-N at Month 0-USA: number analyzed (Participants) | 85 | 67 | 83 | 49 | 42 | 36 | 78 | 77 | 82 | 69 | 71
  CD8+-N-N at Month 0-USA | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+-N-Y at Month 0-Peru: number analyzed (Participants) | 5 | 32 | 0 | 5 | 33 | 33 | 4 | 11 | 7 | 13 | 11
  CD8+-N-Y at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.3 [0.1 to 0.6] |  | 0.3 [0.2 to 0.4] | 0.3 [0.1 to 0.6] | 0.4 [0.2 to 1] | 0.5 [0.5 to 0.6] | 0.6 [0.3 to 5.3] | 0.4 [0.3 to 0.8] | 0.2 [0.1 to 0.6] | 0.4 [0.2 to 0.5]
  CD8+-N-Y at Month 0-Total: number analyzed (Participants) | 12 | 57 | 9 | 48 | 83 | 89 | 18 | 26 | 17 | 36 | 32
  CD8+-N-Y at Month 0-Total | 0.1 [0.1 to 0.3] | 0.3 [0.1 to 0.6] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 1.2] | 0.4 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5]
  CD8+-N-Y at Month 0-USA: number analyzed (Participants) | 7 | 25 | 9 | 43 | 50 | 56 | 14 | 15 | 10 | 23 | 21
  CD8+-N-Y at Month 0-USA | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.8] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6]
  CD8+-ORF3a6-N at Month 0-Peru: number analyzed (Participants) | 46 | 34 | 50 | 47 | 33 | 33 | 48 | 44 | 45 | 46 | 44
  CD8+-ORF3a6-N at Month 0-Peru | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.7] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.8] | 0.1 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6]
  CD8+-ORF3a6-N at Month 0-Total: number analyzed (Participants) | 73 | 52 | 77 | 61 | 44 | 43 | 75 | 68 | 69 | 66 | 66
  CD8+-ORF3a6-N at Month 0-Total | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.5]
  CD8+-ORF3a6-N at Month 0-USA: number analyzed (Participants) | 27 | 18 | 27 | 14 | 11 | 10 | 27 | 24 | 24 | 20 | 22
  CD8+-ORF3a6-N at Month 0-USA | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.5] | 0.1 [0.1 to 0.3] | 0.3 [0.2 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6-Y at Month 0-Peru: number analyzed (Participants) | 4 | 16 | 0 | 3 | 17 | 17 | 2 | 6 | 5 | 4 | 6
  CD8+-ORF3a6-Y at Month 0-Peru | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] |  | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.3 [0.2 to 0.8] | 0.1 [0.1 to 0.1] | 1 [0.7 to 1.3] | 0.3 [0.1 to 0.3] | 0.4 [0.2 to 0.6] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6-Y at Month 0-Total: number analyzed (Participants) | 7 | 28 | 3 | 19 | 36 | 37 | 5 | 12 | 11 | 14 | 14
  CD8+-ORF3a6-Y at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.1] | 0.4 [0.1 to 0.9] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+-ORF3a6-Y at Month 0-USA: number analyzed (Participants) | 3 | 12 | 3 | 16 | 19 | 20 | 3 | 6 | 6 | 10 | 8
  CD8+-ORF3a6-Y at Month 0-USA | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.5] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD8+-ORF7a7b8-N at Month 0-Peru: number analyzed (Participants) | 49 | 35 | 51 | 48 | 34 | 34 | 49 | 44 | 46 | 47 | 46
  CD8+-ORF7a7b8-N at Month 0-Peru | 0.3 [0.1 to 0.8] | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.8] | 0.3 [0.1 to 0.8] | 0.3 [0.1 to 0.9] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.7] | 0.3 [0.1 to 0.8]
  CD8+-ORF7a7b8-N at Month 0-Total: number analyzed (Participants) | 67 | 49 | 71 | 59 | 44 | 38 | 66 | 60 | 59 | 60 | 57
  CD8+-ORF7a7b8-N at Month 0-Total | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.7] | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.5] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.7]
  CD8+-ORF7a7b8-N at Month 0-USA: number analyzed (Participants) | 18 | 14 | 20 | 11 | 10 | 4 | 17 | 16 | 13 | 13 | 11
  CD8+-ORF7a7b8-N at Month 0-USA | 0.1 [0.1 to 0.5] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.5] | 0.1 [0.1 to 0.4]
  CD8+-ORF7a7b8-Y at Month 0-Peru: number analyzed (Participants) | 2 | 16 | 0 | 3 | 17 | 17 | 2 | 7 | 5 | 4 | 5
  CD8+-ORF7a7b8-Y at Month 0-Peru | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] |  | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.9] | 0.1 [0.1 to 0.2] | 1.1 [0.6 to 1.9] | 0.2 [0.2 to 0.3] | 0.5 [0.3 to 0.8] | 0.2 [0.2 to 0.3]
  CD8+-ORF7a7b8-Y at Month 0-Total: number analyzed (Participants) | 4 | 22 | 0 | 12 | 27 | 33 | 5 | 11 | 12 | 11 | 14
  CD8+-ORF7a7b8-Y at Month 0-Total | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.4] |  | 0.1 [0.1 to 0.4] | 0.2 [0.1 to 0.4] | 0.3 [0.1 to 0.6] | 0.1 [0.1 to 0.2] | 0.5 [0.2 to 1.4] | 0.2 [0.1 to 0.4] | 0.3 [0.1 to 0.5] | 0.2 [0.1 to 0.4]
  CD8+-ORF7a7b8-Y at Month 0-USA: number analyzed (Participants) | 2 | 6 | 0 | 9 | 10 | 16 | 3 | 4 | 7 | 7 | 9
  CD8+-ORF7a7b8-Y at Month 0-USA | 0.3 [0.2 to 0.3] | 0.3 [0.1 to 0.6] |  | 0.1 [0.1 to 0.4] | 0.3 [0.1 to 0.5] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.3 [0.1 to 0.5] | 0.1 [0.1 to 0.5] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.5]
  CD8+-S1-N at Month 0-Peru: number analyzed (Participants) | 42 | 33 | 42 | 42 | 33 | 31 | 40 | 39 | 39 | 38 | 38
  CD8+-S1-N at Month 0-Peru | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD8+-S1-N at Month 0-Total: number analyzed (Participants) | 71 | 52 | 69 | 52 | 42 | 42 | 63 | 63 | 65 | 63 | 59
  CD8+-S1-N at Month 0-Total | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S1-N at Month 0-USA: number analyzed (Participants) | 29 | 19 | 27 | 10 | 9 | 11 | 23 | 24 | 26 | 25 | 21
  CD8+-S1-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 0.6] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  CD8+-S1-Y at Month 0-Peru: number analyzed (Participants) | 0 | 9 | 0 | 0 | 9 | 11 | 2 | 3 | 3 | 4 | 4
  CD8+-S1-Y at Month 0-Peru |  | 0.1 [0.1 to 0.3] |  |  | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.4 [0.3 to 0.4] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.6] | 0.1 [0.1 to 0.2]
  CD8+-S1-Y at Month 0-Total: number analyzed (Participants) | 0 | 19 | 2 | 19 | 29 | 29 | 8 | 8 | 6 | 8 | 12
  CD8+-S1-Y at Month 0-Total |  | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0 to 0.1] | 0.2 [0.1 to 0.5] | 0.1 [0.1 to 0.2]
  CD8+-S1-Y at Month 0-USA: number analyzed (Participants) | 0 | 10 | 2 | 19 | 20 | 18 | 6 | 5 | 3 | 4 | 8
  CD8+-S1-Y at Month 0-USA |  | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0 [0 to 0.1] | 0.3 [0.2 to 0.5] | 0.1 [0.1 to 0.2]
  CD8+-S2-N at Month 0-Peru: number analyzed (Participants) | 18 | 14 | 18 | 18 | 14 | 15 | 18 | 18 | 18 | 15 | 18
  CD8+-S2-N at Month 0-Peru | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3]
  CD8+-S2-N at Month 0-Total: number analyzed (Participants) | 30 | 24 | 30 | 27 | 23 | 23 | 28 | 29 | 30 | 26 | 28
  CD8+-S2-N at Month 0-Total | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3]
  CD8+-S2-N at Month 0-USA: number analyzed (Participants) | 12 | 10 | 12 | 9 | 9 | 8 | 10 | 11 | 12 | 11 | 10
  CD8+-S2-N at Month 0-USA | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  CD8+-S2-Y at Month 0-Peru: number analyzed (Participants) | 0 | 4 | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 3 | 0
  CD8+-S2-Y at Month 0-Peru |  | 0.1 [0.1 to 0.2] |  |  | 0.1 [0.1 to 0.2] | 0.9 [0.5 to 1.9] |  |  |  | 0.9 [0.5 to 1.9] |
  CD8+-S2-Y at Month 0-Total: number analyzed (Participants) | 0 | 6 | 0 | 3 | 7 | 7 | 2 | 1 | 0 | 4 | 2
  CD8+-S2-Y at Month 0-Total |  | 0.1 [0.1 to 0.2] |  | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.8] | 0.1 [0.1 to 0.1] | 0.6 [0.6 to 0.6] |  | 0.8 [0.5 to 1.4] | 0.1 [0.1 to 0.1]
  CD8+-S2-Y at Month 0-USA: number analyzed (Participants) | 0 | 2 | 0 | 3 | 3 | 4 | 2 | 1 | 0 | 1 | 2
  CD8+-S2-Y at Month 0-USA |  | 0.4 [0.2 to 0.5] |  | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.6 [0.6 to 0.6] |  | 0.6 [0.6 to 0.6] | 0.1 [0.1 to 0.1]
  CD8+-Spike-N at Month 0-Peru: number analyzed (Participants) | 47 | 37 | 47 | 47 | 37 | 35 | 45 | 44 | 44 | 42 | 43
  CD8+-Spike-N at Month 0-Peru | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3]
  CD8+-Spike-N at Month 0-Total: number analyzed (Participants) | 82 | 61 | 80 | 62 | 51 | 50 | 73 | 73 | 76 | 72 | 70
  CD8+-Spike-N at Month 0-Total | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3]
  CD8+-Spike-N at Month 0-USA: number analyzed (Participants) | 35 | 24 | 33 | 15 | 14 | 15 | 28 | 29 | 32 | 30 | 27
  CD8+-Spike-N at Month 0-USA | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 0.2] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
  CD8+-Spike-Y at Month 0-Peru: number analyzed (Participants) | 0 | 10 | 0 | 0 | 10 | 12 | 2 | 3 | 3 | 5 | 4
  CD8+-Spike-Y at Month 0-Peru |  | 0.2 [0.1 to 0.4] |  |  | 0.2 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.4 [0.3 to 0.4] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 2.7] | 0.1 [0.1 to 0.2]
  CD8+-Spike-Y at Month 0-Total: number analyzed (Participants) | 0 | 21 | 2 | 20 | 31 | 32 | 9 | 9 | 6 | 10 | 12
  CD8+-Spike-Y at Month 0-Total |  | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0 to 0.1] | 0.3 [0.2 to 1] | 0.1 [0.1 to 0.2]
  CD8+-Spike-Y at Month 0-USA: number analyzed (Participants) | 0 | 11 | 2 | 20 | 21 | 20 | 7 | 6 | 3 | 5 | 8
  CD8+-Spike-Y at Month 0-USA |  | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0 to 0.1] | 0.4 [0.3 to 0.7] | 0.2 [0.1 to 0.2]

60. Primary Outcome: SARS-CoV-2-specific Memory B Cell Response Magnitude (B Cell) by Region and Comorbidity Group Among America Cohort
Description: SARS-CoV-2-specific B cell responses and B cell phenotypic data was identified and characterized using fluorescently-labelled recombinant Env proteins (S6P and RBD) in combination with a flow cytometry antibody panel on all available samples from the enrollment visit (V1). The sample will be included in the analysis only if the number of IgD- B cells is equal or greater than 1000 for that sample.
  The table summarized SARS-CoV-2-specific Memory B Cell Response Magnitude by flow cytometry at Visit 1, overall and by region and comorbidity group among America Cohort
Time Frame: Measured at Months 0
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Groups:
- Group 1: Any targeted conditions at enrollment
- Group 2: COPD/emphysema/ asthma
- Group 3: Cigarette smoking - current
- Group 4: Cigarette smoking - ever
- Group 5: Diabetes
- Group 6: HIV
- Group 7: Hypertension
- Group 8: Immune system disorders
- Group 9: Marijuana smoking - current
- Group 10: Marijuana smoking - ever
- Group 11: Smoking - any history
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Group 8 | Group 9 | Group 10 | Group 11
Number analyzed (Participants) | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388 | 388
percentage of cells
  %RBD+ IgA+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %RBD+ IgA+ of Memory B Cells-N-Peru | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %RBD+ IgA+ of Memory B Cells-N-Total | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %RBD+ IgA+ of Memory B Cells-N-USA | 0.01 [0 to 0.03] | 0.00 [0 to 0.03] | 0.00 [0 to 0.03] | 0.00 [0 to 0.03] | 0.00 [0 to 0.03] | 0.00 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03] | 0.00 [0 to 0.04] | 0.00 [0 to 0.04]
  %RBD+ IgA+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %RBD+ IgA+ of Memory B Cells-Y-Peru | 0.02 [0 to 0.05] | 0.05 [0.03 to 0.08] | 0.02 [0 to 0.04] | 0.02 [0 to 0.06] | 0.03 [0.01 to 0.08] | 0.01 [0 to 0.02] | 0.02 [0 to 0.05] | 0.01 [0 to 0.02] |  | 0.03 [0 to 0.03] | 0.02 [0 to 0.06]
  %RBD+ IgA+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %RBD+ IgA+ of Memory B Cells-Y-Total | 0.01 [0 to 0.04] | 0.02 [0 to 0.06] | 0.03 [0 to 0.07] | 0.01 [0 to 0.04] | 0.02 [0 to 0.06] | 0.01 [0 to 0.02] | 0.01 [0 to 0.04] | 0.01 [0 to 0.03] | 0.00 [0 to 0.02] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03]
  %RBD+ IgA+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %RBD+ IgA+ of Memory B Cells-Y-USA | 0.00 [0 to 0.03] | 0.02 [0 to 0.05] | 0.05 [0.01 to 0.08] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.01 [0 to 0.04] | 0.00 [0 to 0.02] | 0.00 [0 to 0.04] | 0.00 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.03]
  %RBD+ IgG+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %RBD+ IgG+ of Memory B Cells-N-Peru | 0.16 [0.08 to 0.31] | 0.15 [0.07 to 0.31] | 0.16 [0.08 to 0.33] | 0.15 [0.07 to 0.3] | 0.15 [0.07 to 0.32] | 0.16 [0.09 to 0.33] | 0.15 [0.08 to 0.31] | 0.16 [0.08 to 0.32] | 0.15 [0.07 to 0.32] | 0.16 [0.08 to 0.32] | 0.15 [0.07 to 0.3]
  %RBD+ IgG+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %RBD+ IgG+ of Memory B Cells-N-Total | 0.15 [0.06 to 0.3] | 0.15 [0.06 to 0.3] | 0.15 [0.06 to 0.31] | 0.15 [0.06 to 0.3] | 0.15 [0.05 to 0.3] | 0.16 [0.06 to 0.31] | 0.15 [0.06 to 0.3] | 0.15 [0.06 to 0.31] | 0.16 [0.06 to 0.31] | 0.16 [0.07 to 0.32] | 0.15 [0.06 to 0.31]
  %RBD+ IgG+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %RBD+ IgG+ of Memory B Cells-N-USA | 0.12 [0.04 to 0.24] | 0.15 [0.05 to 0.29] | 0.15 [0.05 to 0.3] | 0.14 [0.05 to 0.28] | 0.14 [0.04 to 0.28] | 0.15 [0.05 to 0.3] | 0.15 [0.05 to 0.28] | 0.14 [0.05 to 0.28] | 0.16 [0.06 to 0.3] | 0.19 [0.06 to 0.32] | 0.16 [0.03 to 0.31]
  %RBD+ IgG+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %RBD+ IgG+ of Memory B Cells-Y-Peru | 0.13 [0.06 to 0.35] | 0.38 [0.19 to 0.46] | 0.12 [0.08 to 0.18] | 0.18 [0.09 to 0.34] | 0.27 [0.12 to 0.4] | 0.08 [0.05 to 0.16] | 0.14 [0.05 to 0.36] | 0.11 [0.06 to 0.18] |  | 0.10 [0.06 to 0.14] | 0.17 [0.09 to 0.33]
  %RBD+ IgG+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %RBD+ IgG+ of Memory B Cells-Y-Total | 0.15 [0.06 to 0.31] | 0.20 [0.1 to 0.37] | 0.12 [0.04 to 0.22] | 0.20 [0.07 to 0.32] | 0.22 [0.11 to 0.32] | 0.12 [0.04 to 0.25] | 0.15 [0.05 to 0.32] | 0.15 [0.05 to 0.28] | 0.06 [0 to 0.14] | 0.13 [0.05 to 0.25] | 0.15 [0.06 to 0.28]
  %RBD+ IgG+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %RBD+ IgG+ of Memory B Cells-Y-USA | 0.16 [0.05 to 0.3] | 0.17 [0.07 to 0.26] | 0.12 [0 to 0.24] | 0.22 [0.06 to 0.29] | 0.21 [0.1 to 0.3] | 0.15 [0.04 to 0.27] | 0.15 [0.05 to 0.29] | 0.19 [0.04 to 0.28] | 0.06 [0 to 0.14] | 0.13 [0.05 to 0.26] | 0.15 [0.05 to 0.26]
  %RBD+ IgM+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %RBD+ IgM+ of Memory B Cells-N-Peru | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %RBD+ IgM+ of Memory B Cells-N-Total | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %RBD+ IgM+ of Memory B Cells-N-USA | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.03] | 0.00 [0 to 0.02]
  %RBD+ IgM+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %RBD+ IgM+ of Memory B Cells-Y-Peru | 0.00 [0 to 0.01] | 0.00 [0 to 0.14] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.01 [0 to 0.03] | 0.00 [0 to 0] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] |  | 0.00 [0 to 0.01] | 0.00 [0 to 0.01]
  %RBD+ IgM+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %RBD+ IgM+ of Memory B Cells-Y-Total | 0.00 [0 to 0.02] | 0.00 [0 to 0.02] | 0.01 [0 to 0.03] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02]
  %RBD+ IgM+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %RBD+ IgM+ of Memory B Cells-Y-USA | 0.00 [0 to 0.02] | 0.00 [0 to 0.02] | 0.02 [0 to 0.05] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0] | 0.00 [0 to 0.02] | 0.00 [0 to 0.02]
  %RBD+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %RBD+ of Total B Cells-N-Peru | 0.07 [0.05 to 0.12] | 0.08 [0.05 to 0.13] | 0.08 [0.05 to 0.13] | 0.08 [0.05 to 0.13] | 0.07 [0.04 to 0.13] | 0.08 [0.05 to 0.13] | 0.07 [0.05 to 0.12] | 0.08 [0.05 to 0.13] | 0.08 [0.05 to 0.13] | 0.08 [0.05 to 0.13] | 0.08 [0.05 to 0.13]
  %RBD+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %RBD+ of Total B Cells-N-Total | 0.06 [0.03 to 0.11] | 0.07 [0.04 to 0.12] | 0.07 [0.04 to 0.12] | 0.06 [0.03 to 0.12] | 0.06 [0.03 to 0.12] | 0.07 [0.04 to 0.12] | 0.07 [0.04 to 0.11] | 0.07 [0.04 to 0.12] | 0.07 [0.04 to 0.12] | 0.07 [0.04 to 0.13] | 0.07 [0.04 to 0.12]
  %RBD+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %RBD+ of Total B Cells-N-USA | 0.04 [0.02 to 0.07] | 0.05 [0.03 to 0.1] | 0.05 [0.03 to 0.09] | 0.05 [0.03 to 0.09] | 0.05 [0.03 to 0.09] | 0.05 [0.03 to 0.1] | 0.04 [0.03 to 0.09] | 0.05 [0.03 to 0.1] | 0.06 [0.03 to 0.1] | 0.06 [0.03 to 0.12] | 0.04 [0.03 to 0.12]
  %RBD+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %RBD+ of Total B Cells-Y-Peru | 0.10 [0.05 to 0.16] | 0.19 [0.11 to 0.28] | 0.05 [0.04 to 0.07] | 0.08 [0.05 to 0.13] | 0.10 [0.07 to 0.13] | 0.05 [0.04 to 0.12] | 0.12 [0.04 to 0.15] | 0.07 [0.04 to 0.16] |  | 0.07 [0.05 to 0.09] | 0.08 [0.05 to 0.13]
  %RBD+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %RBD+ of Total B Cells-Y-Total | 0.07 [0.04 to 0.13] | 0.06 [0.04 to 0.13] | 0.07 [0.04 to 0.17] | 0.07 [0.04 to 0.12] | 0.08 [0.06 to 0.11] | 0.06 [0.04 to 0.13] | 0.07 [0.04 to 0.13] | 0.06 [0.04 to 0.12] | 0.03 [0.02 to 0.05] | 0.05 [0.03 to 0.09] | 0.06 [0.04 to 0.11]
  %RBD+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %RBD+ of Total B Cells-Y-USA | 0.06 [0.04 to 0.1] | 0.05 [0.03 to 0.11] | 0.14 [0.03 to 0.27] | 0.06 [0.04 to 0.1] | 0.06 [0.05 to 0.1] | 0.06 [0.04 to 0.13] | 0.06 [0.04 to 0.11] | 0.06 [0.03 to 0.09] | 0.03 [0.02 to 0.05] | 0.05 [0.03 to 0.09] | 0.06 [0.03 to 0.09]
  %S+ IgA+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgA+ of Memory B Cells-N-Peru | 0.08 [0.03 to 0.12] | 0.07 [0.03 to 0.12] | 0.07 [0.03 to 0.13] | 0.07 [0.03 to 0.12] | 0.07 [0.03 to 0.12] | 0.08 [0.03 to 0.13] | 0.08 [0.03 to 0.13] | 0.08 [0.03 to 0.13] | 0.07 [0.03 to 0.13] | 0.07 [0.03 to 0.13] | 0.07 [0.03 to 0.12]
  %S+ IgA+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgA+ of Memory B Cells-N-Total | 0.07 [0.03 to 0.11] | 0.06 [0.03 to 0.11] | 0.06 [0.03 to 0.11] | 0.06 [0.03 to 0.11] | 0.06 [0.03 to 0.11] | 0.07 [0.03 to 0.11] | 0.07 [0.03 to 0.11] | 0.07 [0.03 to 0.11] | 0.07 [0.03 to 0.11] | 0.07 [0.03 to 0.12] | 0.06 [0.03 to 0.12]
  %S+ IgA+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgA+ of Memory B Cells-N-USA | 0.06 [0.03 to 0.09] | 0.06 [0.02 to 0.09] | 0.06 [0.02 to 0.1] | 0.06 [0.02 to 0.1] | 0.06 [0.02 to 0.1] | 0.06 [0.02 to 0.1] | 0.06 [0.03 to 0.1] | 0.06 [0.02 to 0.1] | 0.06 [0.02 to 0.1] | 0.06 [0.02 to 0.11] | 0.06 [0.02 to 0.11]
  %S+ IgA+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgA+ of Memory B Cells-Y-Peru | 0.07 [0.03 to 0.13] | 0.14 [0.08 to 0.18] | 0.10 [0.08 to 0.14] | 0.08 [0.03 to 0.13] | 0.14 [0.08 to 0.23] | 0.04 [0.02 to 0.1] | 0.05 [0.01 to 0.11] | 0.05 [0.02 to 0.12] |  | 0.10 [0.06 to 0.12] | 0.08 [0.03 to 0.13]
  %S+ IgA+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgA+ of Memory B Cells-Y-Total | 0.06 [0.02 to 0.11] | 0.07 [0.04 to 0.12] | 0.08 [0.04 to 0.11] | 0.07 [0.03 to 0.11] | 0.08 [0.04 to 0.15] | 0.06 [0.03 to 0.1] | 0.06 [0.01 to 0.1] | 0.06 [0.02 to 0.1] | 0.04 [0.02 to 0.06] | 0.06 [0.02 to 0.09] | 0.07 [0.03 to 0.1]
  %S+ IgA+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgA+ of Memory B Cells-Y-USA | 0.06 [0.02 to 0.1] | 0.06 [0.03 to 0.11] | 0.06 [0.02 to 0.09] | 0.06 [0.03 to 0.09] | 0.07 [0.03 to 0.1] | 0.06 [0.04 to 0.09] | 0.06 [0.01 to 0.1] | 0.06 [0.02 to 0.1] | 0.04 [0.02 to 0.06] | 0.05 [0.02 to 0.08] | 0.06 [0.02 to 0.09]
  %S+ IgA+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgA+ of Total B Cells-N-Peru | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  %S+ IgA+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgA+ of Total B Cells-N-Total | 0.01 [0.01 to 0.03] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.03] | 0.01 [0 to 0.03]
  %S+ IgA+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgA+ of Total B Cells-N-USA | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgA+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgA+ of Total B Cells-Y-Peru | 0.02 [0.01 to 0.04] | 0.03 [0.02 to 0.04] | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04] | 0.04 [0.02 to 0.06] | 0.01 [0.01 to 0.02] | 0.02 [0 to 0.03] | 0.02 [0.01 to 0.03] |  | 0.02 [0.01 to 0.04] | 0.02 [0.01 to 0.04]
  %S+ IgA+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgA+ of Total B Cells-Y-Total | 0.01 [0 to 0.02] | 0.02 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.04] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02]
  %S+ IgA+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgA+ of Total B Cells-Y-USA | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgG+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgG+ of Memory B Cells-N-Peru | 0.79 [0.4 to 1.22] | 0.71 [0.38 to 1.21] | 0.73 [0.41 to 1.22] | 0.64 [0.37 to 1.23] | 0.68 [0.37 to 1.21] | 0.81 [0.42 to 1.23] | 0.75 [0.42 to 1.24] | 0.79 [0.41 to 1.22] | 0.72 [0.39 to 1.22] | 0.77 [0.4 to 1.22] | 0.67 [0.37 to 1.23]
  %S+ IgG+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgG+ of Memory B Cells-N-Total | 0.69 [0.36 to 1.21] | 0.68 [0.33 to 1.2] | 0.72 [0.36 to 1.22] | 0.63 [0.34 to 1.21] | 0.63 [0.31 to 1.2] | 0.72 [0.36 to 1.24] | 0.68 [0.35 to 1.21] | 0.69 [0.36 to 1.22] | 0.71 [0.35 to 1.23] | 0.73 [0.37 to 1.26] | 0.64 [0.36 to 1.22]
  %S+ IgG+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgG+ of Memory B Cells-N-USA | 0.56 [0.32 to 1.11] | 0.67 [0.25 to 1.15] | 0.69 [0.32 to 1.27] | 0.58 [0.31 to 1.06] | 0.57 [0.23 to 1.14] | 0.67 [0.32 to 1.29] | 0.56 [0.3 to 1.07] | 0.63 [0.31 to 1.23] | 0.69 [0.31 to 1.33] | 0.68 [0.31 to 1.43] | 0.61 [0.3 to 1.21]
  %S+ IgG+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgG+ of Memory B Cells-Y-Peru | 0.64 [0.39 to 1.2] | 1.20 [0.83 to 1.53] | 0.47 [0.39 to 0.93] | 0.81 [0.43 to 1.18] | 1.05 [0.62 to 1.23] | 0.52 [0.29 to 0.64] | 0.62 [0.35 to 1.01] | 0.62 [0.4 to 0.86] |  | 0.51 [0.28 to 0.62] | 0.81 [0.43 to 1.17]
  %S+ IgG+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgG+ of Memory B Cells-Y-Total | 0.66 [0.29 to 1.21] | 0.72 [0.31 to 1.53] | 0.29 [0.09 to 0.52] | 0.81 [0.29 to 1.31] | 1.01 [0.57 to 1.27] | 0.50 [0.18 to 0.86] | 0.68 [0.08 to 1.17] | 0.63 [0.24 to 1.08] | 0.29 [0.05 to 0.48] | 0.52 [0.15 to 0.97] | 0.69 [0.29 to 1.15]
  %S+ IgG+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgG+ of Memory B Cells-Y-USA | 0.68 [0.16 to 1.19] | 0.53 [0.25 to 1.28] | 0.16 [0.07 to 0.33] | 0.75 [0.13 to 1.37] | 0.97 [0.55 to 1.27] | 0.36 [0.15 to 0.97] | 0.76 [0.08 to 1.44] | 0.63 [0.16 to 1.12] | 0.29 [0.05 to 0.48] | 0.55 [0.15 to 0.97] | 0.63 [0.16 to 1.12]
  %S+ IgG+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgG+ of Total B Cells-N-Peru | 0.18 [0.09 to 0.25] | 0.18 [0.08 to 0.27] | 0.20 [0.09 to 0.29] | 0.19 [0.09 to 0.29] | 0.18 [0.08 to 0.26] | 0.20 [0.1 to 0.29] | 0.18 [0.08 to 0.27] | 0.19 [0.1 to 0.27] | 0.19 [0.08 to 0.27] | 0.19 [0.09 to 0.29] | 0.19 [0.09 to 0.29]
  %S+ IgG+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgG+ of Total B Cells-N-Total | 0.15 [0.08 to 0.23] | 0.14 [0.06 to 0.24] | 0.15 [0.07 to 0.24] | 0.14 [0.06 to 0.25] | 0.13 [0.06 to 0.23] | 0.15 [0.07 to 0.25] | 0.14 [0.07 to 0.23] | 0.15 [0.07 to 0.25] | 0.15 [0.07 to 0.24] | 0.16 [0.07 to 0.25] | 0.16 [0.07 to 0.25]
  %S+ IgG+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgG+ of Total B Cells-N-USA | 0.10 [0.05 to 0.14] | 0.11 [0.04 to 0.18] | 0.12 [0.05 to 0.19] | 0.11 [0.05 to 0.18] | 0.10 [0.04 to 0.17] | 0.12 [0.04 to 0.18] | 0.10 [0.05 to 0.16] | 0.11 [0.05 to 0.18] | 0.12 [0.05 to 0.19] | 0.12 [0.05 to 0.21] | 0.11 [0.05 to 0.19]
  %S+ IgG+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgG+ of Total B Cells-Y-Peru | 0.19 [0.08 to 0.31] | 0.24 [0.21 to 0.39] | 0.10 [0.08 to 0.16] | 0.19 [0.08 to 0.27] | 0.27 [0.17 to 0.32] | 0.09 [0.06 to 0.19] | 0.19 [0.08 to 0.29] | 0.14 [0.07 to 0.31] |  | 0.15 [0.07 to 0.18] | 0.18 [0.08 to 0.26]
  %S+ IgG+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgG+ of Total B Cells-Y-Total | 0.13 [0.05 to 0.25] | 0.12 [0.05 to 0.24] | 0.06 [0.01 to 0.13] | 0.13 [0.06 to 0.23] | 0.18 [0.12 to 0.28] | 0.09 [0.05 to 0.19] | 0.14 [0.01 to 0.25] | 0.11 [0.05 to 0.22] | 0.04 [0.01 to 0.11] | 0.10 [0.04 to 0.17] | 0.13 [0.06 to 0.21]
  %S+ IgG+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgG+ of Total B Cells-Y-USA | 0.12 [0.04 to 0.21] | 0.11 [0.04 to 0.17] | 0.04 [0 to 0.08] | 0.11 [0.03 to 0.19] | 0.16 [0.11 to 0.24] | 0.08 [0.04 to 0.17] | 0.12 [0.01 to 0.24] | 0.11 [0.04 to 0.19] | 0.04 [0.01 to 0.11] | 0.10 [0.04 to 0.17] | 0.11 [0.04 to 0.17]
  %S+ IgM+ IgD+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgM+ IgD+ of Total B Cells-N-Peru | 0.12 [0.09 to 0.15] | 0.11 [0.08 to 0.15] | 0.11 [0.08 to 0.15] | 0.11 [0.08 to 0.15] | 0.12 [0.08 to 0.15] | 0.12 [0.08 to 0.15] | 0.12 [0.08 to 0.15] | 0.12 [0.08 to 0.15] | 0.12 [0.08 to 0.15] | 0.11 [0.08 to 0.15] | 0.11 [0.08 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgM+ IgD+ of Total B Cells-N-Total | 0.11 [0.08 to 0.15] | 0.10 [0.07 to 0.14] | 0.10 [0.07 to 0.14] | 0.10 [0.08 to 0.14] | 0.10 [0.07 to 0.14] | 0.10 [0.07 to 0.15] | 0.11 [0.08 to 0.15] | 0.11 [0.08 to 0.15] | 0.10 [0.07 to 0.15] | 0.11 [0.08 to 0.15] | 0.10 [0.08 to 0.15]
  %S+ IgM+ IgD+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgM+ IgD+ of Total B Cells-N-USA | 0.10 [0.07 to 0.13] | 0.09 [0.06 to 0.13] | 0.09 [0.07 to 0.13] | 0.09 [0.07 to 0.14] | 0.09 [0.07 to 0.12] | 0.09 [0.07 to 0.14] | 0.10 [0.07 to 0.12] | 0.10 [0.07 to 0.14] | 0.09 [0.07 to 0.14] | 0.10 [0.07 to 0.15] | 0.09 [0.07 to 0.14]
  %S+ IgM+ IgD+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgM+ IgD+ of Total B Cells-Y-Peru | 0.10 [0.07 to 0.15] | 0.16 [0.13 to 0.37] | 0.15 [0.13 to 0.22] | 0.13 [0.07 to 0.16] | 0.10 [0.08 to 0.14] | 0.10 [0.07 to 0.14] | 0.10 [0.05 to 0.13] | 0.10 [0.07 to 0.15] |  | 0.12 [0.06 to 0.14] | 0.13 [0.07 to 0.16]
  %S+ IgM+ IgD+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgM+ IgD+ of Total B Cells-Y-Total | 0.10 [0.07 to 0.14] | 0.10 [0.08 to 0.16] | 0.10 [0.07 to 0.15] | 0.10 [0.07 to 0.15] | 0.09 [0.06 to 0.14] | 0.09 [0.07 to 0.12] | 0.09 [0.06 to 0.13] | 0.08 [0.07 to 0.12] | 0.07 [0.06 to 0.1] | 0.09 [0.07 to 0.12] | 0.10 [0.07 to 0.14]
  %S+ IgM+ IgD+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgM+ IgD+ of Total B Cells-Y-USA | 0.09 [0.07 to 0.12] | 0.09 [0.07 to 0.12] | 0.10 [0.07 to 0.11] | 0.09 [0.06 to 0.12] | 0.08 [0.06 to 0.12] | 0.09 [0.07 to 0.11] | 0.08 [0.06 to 0.13] | 0.08 [0.07 to 0.11] | 0.07 [0.06 to 0.1] | 0.08 [0.07 to 0.11] | 0.09 [0.07 to 0.12]
  %S+ IgM+ of Memory B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgM+ of Memory B Cells-N-Peru | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.02 to 0.08]
  %S+ IgM+ of Memory B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgM+ of Memory B Cells-N-Total | 0.05 [0.02 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.02 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.02 to 0.08] | 0.05 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.02 to 0.08]
  %S+ IgM+ of Memory B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgM+ of Memory B Cells-N-USA | 0.05 [0.02 to 0.06] | 0.04 [0.01 to 0.08] | 0.05 [0.01 to 0.08] | 0.05 [0.02 to 0.08] | 0.04 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.05 [0.01 to 0.08] | 0.05 [0.01 to 0.08] | 0.05 [0.01 to 0.08] | 0.05 [0.01 to 0.08] | 0.05 [0.02 to 0.08]
  %S+ IgM+ of Memory B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgM+ of Memory B Cells-Y-Peru | 0.04 [0.01 to 0.07] | 0.05 [0.03 to 0.11] | 0.07 [0.05 to 0.07] | 0.04 [0.02 to 0.08] | 0.05 [0.02 to 0.08] | 0.02 [0.01 to 0.04] | 0.04 [0.02 to 0.07] | 0.03 [0.02 to 0.05] |  | 0.04 [0.02 to 0.06] | 0.04 [0.02 to 0.07]
  %S+ IgM+ of Memory B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgM+ of Memory B Cells-Y-Total | 0.04 [0.01 to 0.08] | 0.04 [0 to 0.08] | 0.04 [0.01 to 0.06] | 0.04 [0.01 to 0.08] | 0.04 [0.01 to 0.08] | 0.03 [0.01 to 0.06] | 0.04 [0.01 to 0.08] | 0.03 [0.01 to 0.06] | 0.01 [0 to 0.04] | 0.04 [0.01 to 0.07] | 0.04 [0.01 to 0.07]
  %S+ IgM+ of Memory B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgM+ of Memory B Cells-Y-USA | 0.04 [0.01 to 0.08] | 0.04 [0 to 0.07] | 0.02 [0 to 0.05] | 0.04 [0 to 0.07] | 0.02 [0 to 0.08] | 0.03 [0.01 to 0.07] | 0.03 [0 to 0.08] | 0.03 [0.01 to 0.07] | 0.01 [0 to 0.04] | 0.04 [0.01 to 0.07] | 0.04 [0 to 0.07]
  %S+ IgM+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ IgM+ of Total B Cells-N-Peru | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ IgM+ of Total B Cells-N-Total | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ IgM+ of Total B Cells-N-USA | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.01]
  %S+ IgM+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ IgM+ of Total B Cells-Y-Peru | 0.01 [0 to 0.02] | 0.02 [0.01 to 0.02] | 0.01 [0.01 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] |  | 0.01 [0.01 to 0.01] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ IgM+ of Total B Cells-Y-Total | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.00 [0 to 0.02] | 0.01 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.01 [0 to 0.01] | 0.01 [0 to 0.02]
  %S+ IgM+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ IgM+ of Total B Cells-Y-USA | 0.01 [0 to 0.02] | 0.01 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.00 [0 to 0.01] | 0.00 [0 to 0.02] | 0.01 [0 to 0.01] | 0.00 [0 to 0.01] | 0.00 [0 to 0.01] | 0.01 [0 to 0.02] | 0.01 [0 to 0.02]
  %S+ of Total B Cells-N-Peru: number analyzed (Participants) | 88 | 140 | 140 | 103 | 129 | 131 | 124 | 124 | 146 | 139 | 102
  %S+ of Total B Cells-N-Peru | 0.40 [0.29 to 0.52] | 0.40 [0.28 to 0.52] | 0.40 [0.28 to 0.54] | 0.40 [0.28 to 0.54] | 0.39 [0.26 to 0.54] | 0.42 [0.29 to 0.54] | 0.40 [0.28 to 0.55] | 0.40 [0.28 to 0.53] | 0.40 [0.28 to 0.54] | 0.40 [0.28 to 0.54] | 0.40 [0.27 to 0.54]
  %S+ of Total B Cells-N-Total: number analyzed (Participants) | 135 | 263 | 270 | 197 | 251 | 248 | 215 | 224 | 273 | 214 | 162
  %S+ of Total B Cells-N-Total | 0.34 [0.24 to 0.48] | 0.33 [0.21 to 0.49] | 0.33 [0.22 to 0.5] | 0.33 [0.22 to 0.5] | 0.32 [0.2 to 0.49] | 0.34 [0.23 to 0.5] | 0.33 [0.22 to 0.5] | 0.35 [0.23 to 0.5] | 0.34 [0.23 to 0.5] | 0.38 [0.24 to 0.52] | 0.36 [0.23 to 0.52]
  %S+ of Total B Cells-N-USA: number analyzed (Participants) | 47 | 123 | 130 | 94 | 122 | 117 | 91 | 100 | 127 | 75 | 60
  %S+ of Total B Cells-N-USA | 0.26 [0.2 to 0.36] | 0.28 [0.18 to 0.39] | 0.28 [0.2 to 0.4] | 0.28 [0.19 to 0.43] | 0.26 [0.17 to 0.38] | 0.28 [0.19 to 0.41] | 0.26 [0.2 to 0.37] | 0.28 [0.19 to 0.42] | 0.28 [0.2 to 0.42] | 0.30 [0.21 to 0.46] | 0.28 [0.21 to 0.46]
  %S+ of Total B Cells-Y-Peru: number analyzed (Participants) | 58 | 6 | 6 | 43 | 17 | 15 | 22 | 22 | 0 | 7 | 44
  %S+ of Total B Cells-Y-Peru | 0.39 [0.25 to 0.54] | 0.65 [0.44 to 0.99] | 0.37 [0.29 to 0.49] | 0.41 [0.28 to 0.51] | 0.51 [0.36 to 0.71] | 0.29 [0.18 to 0.37] | 0.37 [0.2 to 0.51] | 0.37 [0.23 to 0.63] |  | 0.33 [0.24 to 0.42] | 0.41 [0.29 to 0.51]
  %S+ of Total B Cells-Y-Total: number analyzed (Participants) | 156 | 28 | 21 | 94 | 40 | 43 | 76 | 67 | 18 | 77 | 129
  %S+ of Total B Cells-Y-Total | 0.32 [0.18 to 0.5] | 0.29 [0.21 to 0.53] | 0.26 [0.15 to 0.38] | 0.33 [0.2 to 0.44] | 0.39 [0.29 to 0.52] | 0.28 [0.17 to 0.36] | 0.33 [0.15 to 0.49] | 0.28 [0.17 to 0.41] | 0.19 [0.11 to 0.29] | 0.27 [0.17 to 0.35] | 0.30 [0.18 to 0.42]
  %S+ of Total B Cells-Y-USA: number analyzed (Participants) | 98 | 22 | 15 | 51 | 23 | 28 | 54 | 45 | 18 | 70 | 85
  %S+ of Total B Cells-Y-USA | 0.28 [0.16 to 0.42] | 0.27 [0.19 to 0.48] | 0.15 [0.13 to 0.31] | 0.28 [0.16 to 0.36] | 0.33 [0.25 to 0.46] | 0.26 [0.17 to 0.35] | 0.29 [0.15 to 0.48] | 0.25 [0.15 to 0.34] | 0.19 [0.11 to 0.29] | 0.26 [0.17 to 0.35] | 0.28 [0.17 to 0.36]

61. Primary Outcome: SARS-CoV-2-specific Infection Presentation, Including Clinical Course, Along With Demographics and Corresponding Medical History of Participants , Overall and by Region Among America Cohort
Description: SARS-CoV-2-specific Infection Presentation, Including Clinical Course, Along With Demographics and Corresponding Medical History of Participants , overall and by region
Time Frame: Measured at Months 0
Population: American Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
Participants
  Any targeted conditions at enrollment | 14 | 21 | 18 | 32 | 20 | 33 | 53
  COPD/emphysema/ asthma | 2 | 23 | 6 | 6 | 4 | 8 | 11
  Chronic kidney disease | 0 | 28 | 0 | 0 | 0 | 1 | 2
  Cigarette smoking - current | 5 | 18 | 4 | 1 | 2 | 0 | 9
  Cigarette smoking - ever | 11 | 17 | 15 | 19 | 11 | 18 | 37
  Congestive heart failure | 0 | 24 | 0 | 0 | 1 | 3 | 3
  Currently smoke cigarettes or marijua0 | 8 | 5 | 8 | 2 | 3 | 2 | 12
  Diabetes | 3 | 26 | 3 | 8 | 7 | 9 | 12
  Diabetes with complications | 1 | 27 | 0 | 1 | 1 | 0 | 3
  Ever smoked cigarettes or marijua0 | 18 | 16 | 23 | 25 | 15 | 24 | 47
  HIV | 4 | 29 | 6 | 2 | 4 | 4 | 21
  Hypertension | 6 | 22 | 2 | 20 | 12 | 17 | 22
  Immune system disorders | 5 | 30 | 11 | 6 | 6 | 14 | 29
  Immune system disorders, non HIV | 1 | 31 | 5 | 4 | 2 | 10 | 8
  Marijua0 smoking - current | 4 | 20 | 4 | 1 | 2 | 2 | 6
  Marijua0 smoking - ever | 11 | 19 | 17 | 14 | 7 | 17 | 26
  Myocarditis/ pericarditis | 0 | 25 | 0 | 0 | 0 | 0 | 1
  Prolonged viral shedding | 1 | 0 | 3 | 2 | 0 | 0 | 30

62. Primary Outcome: SARS-CoV-2-specific Infection Presentation, Including Clinical Course, Along With Demographics and Corresponding Medical History of Participants , Overall and by Region Among Africa Cohort
Description: as for outcome 61
Time Frame: Measured at Months 0
Population: african Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 79 | 17 | 129 | 26 | 73 | 24 | 24
Participants
  Any targeted conditions at enrollment | 14 | 12 | 44 | 17 | 38 | 20 | 13
  COPD/emphysema/ asthma | 0 | 2 | 9 | 0 | 2 | 1 | 3
  Chronic kidney disease | 1 | 0 | 0 | 1 | 2 | 2 | 0
  Congestive heart failure | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Currently smoke cigarettes or marijua0 | 12 | 1 | 12 | 3 | 4 | 2 | 2
  Diabetes | 4 | 3 | 11 | 6 | 15 | 10 | 4
  Diabetes with complications | 1 | 0 | 0 | 1 | 2 | 2 | 1
  Ever smoked cigarettes or marijua0 | 20 | 2 | 27 | 6 | 10 | 4 | 6
  HIV | 6 | 2 | 14 | 0 | 18 | 2 | 2
  Hypertension | 7 | 8 | 15 | 15 | 18 | 18 | 8
  Immune system disorders | 6 | 2 | 15 | 0 | 18 | 3 | 3
  Immune system disorders, non HIV | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Myocarditis/ pericarditis | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Prolonged viral shedding | 1 | 0 | 2 | 0 | 1 | 0 | 1

63. Secondary Outcome: SARS-CoV-2-specific Antibody Binding Response Magnitude (IgA Nasal Sample) by Region and Enrollment Group Among America Cohort
Description: BAMA assays was performed for samples from participants at Visit 1 (Month 0, baseline) and available samples at follow-up visits (Month 2, 4). Serum SARS-CoV-2-specific IgA, IgG1, IgG3 responses (dilution 1:50) to SARS-CoV-2 antigens were measured on a Bio-Plex instrument (Bio-Rad). The Bioplex software provides 2 readouts: a background-subtracted mean fluorescence intensity (MFI), where background refers to a plate level control (i.e., a blank well run on each plate), and a concentration based on a standard curve. Positive responses at each visit will be called if the MFI minus blank values are ≥ isotype, antigen, and dilution-specific cutoff (will be provided by the lab). MFIs minus blank (or net MFI) are used to summarize the magnitude at a given time-point.
  The table summarized SARS-CoV-2-specific Antibody Binding Response Magnitude by binding antibody multiplex assay (BAMA IgA nasal sample) at Visit 1, 2, 3, overall and by region and enrollment group among America Cohort
Time Frame: Measured at Months 0, 2, 5
Population: American Population (USA and Peru only), all available data at each visit
Measure: Median (Inter-Quartile Range); unit: MFI
Groups:
- Group 1A: Asymptomatic, age 18 - 55
- Group 1B: Asymptomatic, age 55+
- Group 1C: Symptomatic, age 18 - 55
- Group 1D: Symptomatic, age 55+
- Group 2A: Hospitalized, age 18 - 55
- Group 2B: Hospitalized, age 55+
- Group 3: Clinical spectrums
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 50 | 34 | 53 | 51 | 49 | 50 | 101
MFI
  2019-nCoV S/293F at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  2019-nCoV S/293F at Month 0-Peru |  | 1.88 [1.88 to 1.88] |  |  |  |  |
  2019-nCoV S/293F at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  2019-nCoV S/293F at Month 0-Total | 2.67 [2.24 to 3.1] | 1.36 [0.72 to 1.62] | 0.2 [0.09 to 0.28] | 0.41 [0.12 to 2.02] | 1.13 [0.91 to 1.36] | 0.55 [0.38 to 1.86] | 0.88 [0.18 to 2.26]
  2019-nCoV S/293F at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  2019-nCoV S/293F at Month 0-USA | 2.67 [2.24 to 3.1] | 0.72 [0.41 to 1.04] | 0.2 [0.09 to 0.28] | 0.41 [0.12 to 2.02] | 1.13 [0.91 to 1.36] | 0.55 [0.38 to 1.86] | 0.88 [0.18 to 2.26]
  2019-nCoV S/293F at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  2019-nCoV S/293F at Month 2-Peru | 0.32 [0.18 to 0.94] | 0.1 [0.1 to 0.1] | 0.51 [0.17 to 0.65] | 0.09 [0.09 to 0.35] | 1.98 [0.64 to 3.8] | 10.13 [10.13 to 10.13] | 1.78 [1.22 to 2.09]
  2019-nCoV S/293F at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  2019-nCoV S/293F at Month 2-Total | 0.46 [0.2 to 1.07] | 0.1 [0.09 to 0.1] | 0.56 [0.17 to 0.84] | 0.75 [0.18 to 2.72] | 0.67 [0.51 to 3.63] | 4.8 [2.47 to 7.46] | 1 [0.63 to 2.19]
  2019-nCoV S/293F at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  2019-nCoV S/293F at Month 2-USA | 2.25 [2.25 to 2.25] | 0.09 [0.09 to 0.09] | 0.58 [0.13 to 0.95] | 2.32 [0.57 to 2.73] | 0.38 [0.38 to 0.38] | 2.47 [1.3 to 3.63] | 1 [0.47 to 1.68]
  2019-nCoV S/293F at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  2019-nCoV S/293F at Month 4-Peru | 0.16 [0.09 to 0.81] | 0.09 [0.09 to 0.09] | 0.09 [0.09 to 0.11] | 0.62 [0.38 to 0.86] | 0.72 [0.17 to 2.66] | 1.53 [1.38 to 1.67] | 4 [1.66 to 4.18]
  2019-nCoV S/293F at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  2019-nCoV S/293F at Month 4-Total | 0.16 [0.09 to 0.81] | 0.09 [0.09 to 0.09] | 0.12 [0.09 to 0.37] | 0.89 [0.22 to 1.25] | 0.72 [0.17 to 2.66] | 1.46 [1.22 to 1.71] | 0.74 [0.5 to 4.09]
  2019-nCoV S/293F at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  2019-nCoV S/293F at Month 4-USA |  |  | 0.46 [0.24 to 2.21] | 0.89 [0.3 to 1.41] |  | 1.42 [1.29 to 1.55] | 0.52 [0.38 to 0.69]
  229E-RBD at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  229E-RBD at Month 0-Peru |  | 0.3 [0.3 to 0.3] |  |  |  |  |
  229E-RBD at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 18
  229E-RBD at Month 0-Total | 0.97 [0.59 to 1.36] | 0.3 [0.15 to 0.55] | 0.4 [0.13 to 1.06] | 1.17 [0.33 to 2.36] | 0.07 [0.06 to 0.08] | 0.54 [0.36 to 1.07] | 0.44 [0.18 to 1.96]
  229E-RBD at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 18
  229E-RBD at Month 0-USA | 0.97 [0.59 to 1.36] | 0.4 [0.2 to 0.6] | 0.4 [0.13 to 1.06] | 1.17 [0.33 to 2.36] | 0.07 [0.06 to 0.08] | 0.54 [0.36 to 1.07] | 0.44 [0.18 to 1.96]
  229E-RBD at Month 2-Peru: number analyzed (Participants) | 12 | 1 | 7 | 3 | 6 | 1 | 3
  229E-RBD at Month 2-Peru | 0.5 [0.44 to 1.74] | 2.75 [2.75 to 2.75] | 0.69 [0.35 to 1.22] | 1.16 [0.67 to 5.86] | 0.58 [0.41 to 0.63] | 5.04 [5.04 to 5.04] | 0.24 [0.18 to 0.31]
  229E-RBD at Month 2-Total: number analyzed (Participants) | 13 | 2 | 18 | 14 | 7 | 3 | 13
  229E-RBD at Month 2-Total | 0.5 [0.45 to 1.64] | 1.72 [1.21 to 2.23] | 0.59 [0.18 to 1.07] | 1.66 [0.6 to 3.05] | 0.54 [0.33 to 0.62] | 1 [0.82 to 3.02] | 0.31 [0.12 to 1.87]
  229E-RBD at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 10
  229E-RBD at Month 2-USA | 1.64 [1.64 to 1.64] | 0.7 [0.7 to 0.7] | 0.49 [0.13 to 1] | 1.66 [0.67 to 2.73] | 0.28 [0.28 to 0.28] | 0.82 [0.74 to 0.91] | 0.59 [0.11 to 2.32]
  229E-RBD at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  229E-RBD at Month 4-Peru | 0.48 [0.32 to 1.17] | 2.63 [2.63 to 2.63] | 0.25 [0.22 to 0.57] | 1.84 [1.25 to 2.43] | 0.29 [0.2 to 0.38] | 6.17 [3.48 to 8.86] | 0.55 [0.38 to 1.57]
  229E-RBD at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  229E-RBD at Month 4-Total | 0.48 [0.32 to 1.17] | 2.63 [2.63 to 2.63] | 0.25 [0.15 to 0.85] | 1.92 [0.45 to 2.91] | 0.29 [0.2 to 0.38] | 0.75 [0.58 to 3.48] | 0.55 [0.21 to 1.99]
  229E-RBD at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  229E-RBD at Month 4-USA |  |  | 0.37 [0.09 to 0.94] | 1.92 [0.24 to 2.8] |  | 0.45 [0.32 to 0.58] | 0.72 [0.21 to 2.11]
  HCoV-229E S1S2 ECD His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HCoV-229E S1S2 ECD His at Month 0-Peru |  | 0.7 [0.7 to 0.7] |  |  |  |  |
  HCoV-229E S1S2 ECD His at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  HCoV-229E S1S2 ECD His at Month 0-Total | 0.93 [0.51 to 1.34] | 0.7 [0.67 to 0.79] | 0.69 [0.24 to 1.98] | 1.88 [0.51 to 4.13] | 0.03 [0.02 to 0.03] | 0.74 [0.68 to 1.39] | 1.09 [0.2 to 2.85]
  HCoV-229E S1S2 ECD His at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  HCoV-229E S1S2 ECD His at Month 0-USA | 0.93 [0.51 to 1.34] | 0.77 [0.71 to 0.83] | 0.69 [0.24 to 1.98] | 1.88 [0.51 to 4.13] | 0.03 [0.02 to 0.03] | 0.74 [0.68 to 1.39] | 1.09 [0.2 to 2.85]
  HCoV-229E S1S2 ECD His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  HCoV-229E S1S2 ECD His at Month 2-Peru | 1.36 [0.58 to 3.34] | 2.8 [2.8 to 2.8] | 1.51 [1.39 to 2.57] | 3.32 [1.71 to 6.49] | 1.55 [0.37 to 2.69] | 4.34 [4.34 to 4.34] | 0.67 [0.5 to 1.32]
  HCoV-229E S1S2 ECD His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  HCoV-229E S1S2 ECD His at Month 2-Total | 1.63 [0.66 to 3.22] | 1.7 [1.16 to 2.25] | 1.48 [0.25 to 2.2] | 3.35 [1.56 to 4.64] | 0.64 [0.35 to 2.61] | 1.71 [0.92 to 3.03] | 1.27 [0.34 to 1.98]
  HCoV-229E S1S2 ECD His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  HCoV-229E S1S2 ECD His at Month 2-USA | 1.9 [1.9 to 1.9] | 0.61 [0.61 to 0.61] | 0.42 [0.16 to 2.04] | 3.37 [1.62 to 4.52] | 0.42 [0.42 to 0.42] | 0.92 [0.52 to 1.32] | 1.87 [0.3 to 2.93]
  HCoV-229E S1S2 ECD His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  HCoV-229E S1S2 ECD His at Month 4-Peru | 1.19 [0.49 to 3.09] | 2.79 [2.79 to 2.79] | 2.28 [1.21 to 3.57] | 1.3 [0.98 to 1.63] | 0.45 [0.29 to 1.95] | 3.65 [2.12 to 5.17] | 0.85 [0.83 to 4.43]
  HCoV-229E S1S2 ECD His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  HCoV-229E S1S2 ECD His at Month 4-Total | 1.19 [0.49 to 3.09] | 2.79 [2.79 to 2.79] | 0.98 [0.16 to 1.91] | 1.86 [0.41 to 2.92] | 0.45 [0.29 to 1.95] | 1.28 [0.47 to 3.16] | 0.85 [0.61 to 3.8]
  HCoV-229E S1S2 ECD His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  HCoV-229E S1S2 ECD His at Month 4-USA |  |  | 0.28 [0.1 to 0.71] | 1.86 [0.16 to 3.88] |  | 1.04 [0.57 to 1.51] | 1.34 [0.25 to 2.94]
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-Peru |  | 0.28 [0.28 to 0.28] |  |  |  |  |
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-Total | 2.26 [2.09 to 2.43] | 0.28 [0.19 to 0.45] | 0.12 [0.07 to 1.13] | 0.66 [0.36 to 2.34] | 0.44 [0.3 to 0.58] | 0.81 [0.19 to 2.08] | 0.87 [0.27 to 3.75]
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  HCoV-HKU1 N5 S1S2 ECD His at Month 0-USA | 2.26 [2.09 to 2.43] | 0.37 [0.23 to 0.5] | 0.12 [0.07 to 1.13] | 0.66 [0.36 to 2.34] | 0.44 [0.3 to 0.58] | 0.81 [0.19 to 2.08] | 0.87 [0.27 to 3.75]
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-Peru | 0.72 [0.14 to 1.47] | 0.37 [0.37 to 0.37] | 0.31 [0.28 to 1.1] | 0.48 [0.27 to 1.72] | 2.16 [0.67 to 3.37] | 7.26 [7.26 to 7.26] | 1.17 [0.84 to 2.17]
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-Total | 0.77 [0.15 to 1.61] | 0.23 [0.16 to 0.3] | 0.3 [0.16 to 1.21] | 2.04 [0.35 to 4.5] | 1.42 [0.37 to 3.21] | 2.24 [1.26 to 4.75] | 1.69 [0.64 to 3.11]
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  HCoV-HKU1 N5 S1S2 ECD His at Month 2-USA | 1.66 [1.66 to 1.66] | 0.09 [0.09 to 0.09] | 0.29 [0.1 to 1.24] | 2.34 [0.39 to 5.02] | 0.12 [0.12 to 0.12] | 1.26 [0.77 to 1.75] | 1.72 [0.73 to 3.41]
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-Peru | 0.36 [0.14 to 1.73] | 0.26 [0.26 to 0.26] | 0.2 [0.14 to 0.37] | 0.47 [0.46 to 0.49] | 0.45 [0.2 to 2.47] | 0.75 [0.55 to 0.96] | 2.09 [1.63 to 5.21]
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-Total | 0.36 [0.14 to 1.73] | 0.26 [0.26 to 0.26] | 0.2 [0.14 to 0.68] | 0.5 [0.44 to 0.68] | 0.45 [0.2 to 2.47] | 0.75 [0.3 to 1.51] | 1.95 [0.95 to 3.61]
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  HCoV-HKU1 N5 S1S2 ECD His at Month 4-USA |  |  | 0.39 [0.14 to 1] | 0.51 [0.44 to 0.85] |  | 1.38 [0.78 to 1.97] | 1.33 [0.37 to 2.64]
  HCoV-NL63 S1S2 ECD His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HCoV-NL63 S1S2 ECD His at Month 0-Peru |  | 0.05 [0.05 to 0.05] |  |  |  |  |
  HCoV-NL63 S1S2 ECD His at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  HCoV-NL63 S1S2 ECD His at Month 0-Total | 0.14 [0.12 to 0.16] | 0.05 [0.03 to 0.05] | 0.03 [0.02 to 0.2] | 0.06 [0.03 to 0.15] | 0.06 [0.05 to 0.07] | 0.23 [0.03 to 0.29] | 0.21 [0.03 to 0.28]
  HCoV-NL63 S1S2 ECD His at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  HCoV-NL63 S1S2 ECD His at Month 0-USA | 0.14 [0.12 to 0.16] | 0.03 [0.01 to 0.04] | 0.03 [0.02 to 0.2] | 0.06 [0.03 to 0.15] | 0.06 [0.05 to 0.07] | 0.23 [0.03 to 0.29] | 0.21 [0.03 to 0.28]
  HCoV-NL63 S1S2 ECD His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  HCoV-NL63 S1S2 ECD His at Month 2-Peru | 0.16 [0.08 to 0.39] | 0.11 [0.11 to 0.11] | 0.13 [0.07 to 0.26] | 0.14 [0.09 to 0.72] | 0.57 [0.2 to 1.04] | 0.55 [0.55 to 0.55] | 0.07 [0.06 to 0.33]
  HCoV-NL63 S1S2 ECD His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  HCoV-NL63 S1S2 ECD His at Month 2-Total | 0.19 [0.09 to 0.37] | 0.08 [0.07 to 0.09] | 0.09 [0.04 to 0.28] | 0.22 [0.15 to 0.86] | 0.25 [0.17 to 1] | 0.47 [0.26 to 0.51] | 0.2 [0.08 to 0.44]
  HCoV-NL63 S1S2 ECD His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  HCoV-NL63 S1S2 ECD His at Month 2-USA | 0.23 [0.23 to 0.23] | 0.05 [0.05 to 0.05] | 0.08 [0.02 to 0.23] | 0.27 [0.15 to 0.82] | 0.15 [0.15 to 0.15] | 0.26 [0.15 to 0.37] | 0.21 [0.11 to 0.44]
  HCoV-NL63 S1S2 ECD His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  HCoV-NL63 S1S2 ECD His at Month 4-Peru | 0.09 [0.05 to 0.16] | 0.08 [0.08 to 0.08] | 0.11 [0.05 to 0.26] | 0.18 [0.16 to 0.19] | 0.24 [0.12 to 0.35] | 0.17 [0.1 to 0.24] | 0.15 [0.06 to 0.54]
  HCoV-NL63 S1S2 ECD His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  HCoV-NL63 S1S2 ECD His at Month 4-Total | 0.09 [0.05 to 0.16] | 0.08 [0.08 to 0.08] | 0.05 [0.01 to 0.17] | 0.16 [0.1 to 0.28] | 0.24 [0.12 to 0.35] | 0.17 [0.03 to 0.33] | 0.15 [0.06 to 0.45]
  HCoV-NL63 S1S2 ECD His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  HCoV-NL63 S1S2 ECD His at Month 4-USA |  |  | 0.02 [0.005 to 0.08] | 0.16 [0.06 to 0.34] |  | 0.22 [0.12 to 0.31] | 0.19 [0.07 to 0.35]
  HCoV-OC43 S1S2 ECD His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HCoV-OC43 S1S2 ECD His at Month 0-Peru |  | 0.95 [0.95 to 0.95] |  |  |  |  |
  HCoV-OC43 S1S2 ECD His at Month 0-Total: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  HCoV-OC43 S1S2 ECD His at Month 0-Total | 4.66 [3.77 to 5.54] | 0.74 [0.64 to 0.85] | 0.51 [0.15 to 1.98] | 1.55 [0.66 to 4.23] | 1.05 [0.93 to 1.16] | 1.47 [0.64 to 3.63] | 2.05 [0.8 to 6.71]
  HCoV-OC43 S1S2 ECD His at Month 0-USA: number analyzed (Participants) | 2 | 1 | 11 | 15 | 2 | 5 | 19
  HCoV-OC43 S1S2 ECD His at Month 0-USA | 4.66 [3.77 to 5.54] | 0.53 [0.53 to 0.53] | 0.51 [0.15 to 1.98] | 1.55 [0.66 to 4.23] | 1.05 [0.93 to 1.16] | 1.47 [0.64 to 3.63] | 2.05 [0.8 to 6.71]
  HCoV-OC43 S1S2 ECD His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  HCoV-OC43 S1S2 ECD His at Month 2-Peru | 1.7 [0.56 to 2.99] | 2.23 [2.23 to 2.23] | 1.08 [0.86 to 2.62] | 1.63 [0.86 to 2.18] | 3.22 [1.6 to 5.18] | 7.58 [7.58 to 7.58] | 2.61 [1.76 to 2.62]
  HCoV-OC43 S1S2 ECD His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  HCoV-OC43 S1S2 ECD His at Month 2-Total | 2.07 [0.65 to 4.07] | 1.34 [0.89 to 1.78] | 1.06 [0.48 to 2.71] | 3.02 [0.74 to 5.02] | 2.84 [1.14 to 4.66] | 3.2 [2.05 to 5.39] | 2.99 [1.06 to 6.9]
  HCoV-OC43 S1S2 ECD His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  HCoV-OC43 S1S2 ECD His at Month 2-USA | 4.43 [4.43 to 4.43] | 0.45 [0.45 to 0.45] | 1.02 [0.41 to 2.48] | 3.96 [0.89 to 5.13] | 0.95 [0.95 to 0.95] | 2.05 [1.47 to 2.62] | 4.51 [1.07 to 8.16]
  HCoV-OC43 S1S2 ECD His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  HCoV-OC43 S1S2 ECD His at Month 4-Peru | 1 [0.44 to 4.27] | 1.46 [1.46 to 1.46] | 0.76 [0.32 to 1.32] | 0.59 [0.55 to 0.64] | 1.08 [0.82 to 2.62] | 1.17 [1.02 to 1.32] | 4.38 [3.53 to 6.23]
  HCoV-OC43 S1S2 ECD His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  HCoV-OC43 S1S2 ECD His at Month 4-Total | 1 [0.44 to 4.27] | 1.46 [1.46 to 1.46] | 0.76 [0.3 to 1.96] | 0.77 [0.59 to 1.48] | 1.08 [0.82 to 2.62] | 1.17 [0.79 to 2.66] | 3.53 [1.53 to 5.41]
  HCoV-OC43 S1S2 ECD His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  HCoV-OC43 S1S2 ECD His at Month 4-USA |  |  | 1.23 [0.3 to 3.79] | 1.18 [0.77 to 1.77] |  | 3.4 [1.99 to 4.82] | 2.24 [0.5 to 4.25]
  HKU1-RBD at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HKU1-RBD at Month 0-Peru |  | 0.2 [0.2 to 0.2] |  |  |  |  |
  HKU1-RBD at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  HKU1-RBD at Month 0-Total | 0.85 [0.51 to 1.2] | 0.02 [0.01 to 0.11] | 0.07 [0.04 to 0.55] | 0.29 [0.19 to 0.42] | 0.39 [0.24 to 0.53] | 0.33 [0.21 to 0.76] | 0.17 [0.06 to 0.62]
  HKU1-RBD at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  HKU1-RBD at Month 0-USA | 0.85 [0.51 to 1.2] | 0.01 [0.01 to 0.02] | 0.07 [0.04 to 0.55] | 0.29 [0.19 to 0.42] | 0.39 [0.24 to 0.53] | 0.33 [0.21 to 0.76] | 0.17 [0.06 to 0.62]
  HKU1-RBD at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 2 | 6 | 1 | 3
  HKU1-RBD at Month 2-Peru | 0.28 [0.07 to 0.48] | 0.24 [0.24 to 0.24] | 0.11 [0.04 to 0.22] | 0.09 [0.05 to 0.12] | 0.31 [0.12 to 0.51] | 6.99 [6.99 to 6.99] | 0.51 [0.28 to 1.07]
  HKU1-RBD at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 13 | 7 | 3 | 13
  HKU1-RBD at Month 2-Total | 0.24 [0.09 to 0.48] | 0.13 [0.08 to 0.18] | 0.11 [0.04 to 0.43] | 0.27 [0.15 to 0.51] | 0.15 [0.12 to 0.5] | 0.98 [0.75 to 3.98] | 0.27 [0.1 to 0.69]
  HKU1-RBD at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 10
  HKU1-RBD at Month 2-USA | 0.16 [0.16 to 0.16] | 0.03 [0.03 to 0.03] | 0.11 [0.04 to 0.55] | 0.46 [0.19 to 0.51] | 0.15 [0.15 to 0.15] | 0.75 [0.64 to 0.86] | 0.27 [0.13 to 0.62]
  HKU1-RBD at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  HKU1-RBD at Month 4-Peru | 0.23 [0.05 to 0.72] | 0.21 [0.21 to 0.21] | 0.03 [0.02 to 0.05] | 0.14 [0.13 to 0.15] | 0.11 [0.07 to 0.34] | 1.19 [0.8 to 1.58] | 0.7 [0.64 to 0.81]
  HKU1-RBD at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  HKU1-RBD at Month 4-Total | 0.23 [0.05 to 0.72] | 0.21 [0.21 to 0.21] | 0.07 [0.02 to 0.13] | 0.16 [0.16 to 0.38] | 0.11 [0.07 to 0.34] | 0.64 [0.34 to 1.15] | 0.51 [0.13 to 0.75]
  HKU1-RBD at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  HKU1-RBD at Month 4-USA |  |  | 0.14 [0.08 to 0.21] | 0.32 [0.16 to 0.44] |  | 0.51 [0.33 to 0.69] | 0.27 [0.09 to 0.47]
  NL63-RBD at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NL63-RBD at Month 0-Peru |  | 0.4 [0.4 to 0.4] |  |  |  |  |
  NL63-RBD at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  NL63-RBD at Month 0-Total | 1.65 [1.59 to 1.72] | 0.53 [0.47 to 0.7] | 0.47 [0.21 to 1.75] | 1.27 [0.44 to 2.29] | 0.56 [0.51 to 0.62] | 1.18 [0.28 to 2.34] | 1.11 [0.32 to 1.45]
  NL63-RBD at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  NL63-RBD at Month 0-USA | 1.65 [1.59 to 1.72] | 0.7 [0.61 to 0.78] | 0.47 [0.21 to 1.75] | 1.27 [0.44 to 2.29] | 0.56 [0.51 to 0.62] | 1.18 [0.28 to 2.34] | 1.11 [0.32 to 1.45]
  NL63-RBD at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  NL63-RBD at Month 2-Peru | 0.67 [0.45 to 3.71] | 1.78 [1.78 to 1.78] | 0.76 [0.44 to 2.66] | 2.11 [1.27 to 5.49] | 2.22 [1.44 to 3.69] | 2.67 [2.67 to 2.67] | 0.31 [0.23 to 0.51]
  NL63-RBD at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  NL63-RBD at Month 2-Total | 0.68 [0.48 to 3.2] | 1.36 [1.14 to 1.57] | 0.62 [0.37 to 1.49] | 1.99 [1.2 to 4.25] | 2.05 [1.52 to 3.26] | 1.04 [0.75 to 1.85] | 0.95 [0.25 to 2.09]
  NL63-RBD at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  NL63-RBD at Month 2-USA | 1.66 [1.66 to 1.66] | 0.93 [0.93 to 0.93] | 0.42 [0.21 to 1.13] | 1.87 [1.38 to 3.83] | 1.8 [1.8 to 1.8] | 0.75 [0.61 to 0.89] | 1.1 [0.54 to 3.39]
  NL63-RBD at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  NL63-RBD at Month 4-Peru | 0.87 [0.33 to 3.17] | 2.11 [2.11 to 2.11] | 0.52 [0.34 to 0.79] | 2.24 [2.13 to 2.36] | 1.8 [1.14 to 2.41] | 1.49 [1.03 to 1.94] | 1.49 [0.6 to 2.42]
  NL63-RBD at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  NL63-RBD at Month 4-Total | 0.87 [0.33 to 3.17] | 2.11 [2.11 to 2.11] | 0.46 [0.25 to 0.79] | 2.01 [1.18 to 3.35] | 1.8 [1.14 to 2.41] | 1.3 [0.49 to 2.11] | 1.57 [0.57 to 4.56]
  NL63-RBD at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  NL63-RBD at Month 4-USA |  |  | 0.31 [0.06 to 1.39] | 1.43 [0.93 to 4.23] |  | 1.14 [0.7 to 1.58] | 2.28 [0.8 to 5.35]
  OC43-RBD at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  OC43-RBD at Month 0-Peru |  | 0.36 [0.36 to 0.36] |  |  |  |  |
  OC43-RBD at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  OC43-RBD at Month 0-Total | 0.86 [0.71 to 1] | 0.17 [0.08 to 0.26] | 0.2 [0.03 to 0.39] | 0.19 [0.15 to 0.74] | 0.52 [0.37 to 0.67] | 0.46 [0.36 to 0.48] | 0.2 [0.11 to 0.51]
  OC43-RBD at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  OC43-RBD at Month 0-USA | 0.86 [0.71 to 1] | 0.08 [0.04 to 0.13] | 0.2 [0.03 to 0.39] | 0.19 [0.15 to 0.74] | 0.52 [0.37 to 0.67] | 0.46 [0.36 to 0.48] | 0.2 [0.11 to 0.51]
  OC43-RBD at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 5 | 1 | 3
  OC43-RBD at Month 2-Peru | 0.18 [0.08 to 0.85] | 1.27 [1.27 to 1.27] | 0.13 [0.05 to 0.21] | 0.97 [0.5 to 1.38] | 0.19 [0.14 to 0.33] | 3.44 [3.44 to 3.44] | 0.25 [0.18 to 0.27]
  OC43-RBD at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 6 | 3 | 13
  OC43-RBD at Month 2-Total | 0.4 [0.09 to 0.99] | 0.7 [0.41 to 0.98] | 0.11 [0.05 to 0.39] | 0.7 [0.31 to 1.21] | 0.26 [0.15 to 0.33] | 1.71 [1.16 to 2.57] | 0.19 [0.11 to 0.3]
  OC43-RBD at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 10
  OC43-RBD at Month 2-USA | 1.04 [1.04 to 1.04] | 0.13 [0.13 to 0.13] | 0.09 [0.05 to 0.44] | 0.44 [0.31 to 1.15] | 0.33 [0.33 to 0.33] | 1.16 [0.89 to 1.43] | 0.16 [0.11 to 0.54]
  OC43-RBD at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  OC43-RBD at Month 4-Peru | 0.12 [0.08 to 0.76] | 1.09 [1.09 to 1.09] | 0.06 [0.02 to 0.11] | 0.25 [0.2 to 0.3] | 0.1 [0.06 to 0.27] | 0.65 [0.6 to 0.7] | 0.44 [0.38 to 0.84]
  OC43-RBD at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  OC43-RBD at Month 4-Total | 0.12 [0.08 to 0.76] | 1.09 [1.09 to 1.09] | 0.07 [0.02 to 0.15] | 0.38 [0.25 to 0.53] | 0.1 [0.06 to 0.27] | 0.52 [0.41 to 0.6] | 0.38 [0.09 to 0.64]
  OC43-RBD at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  OC43-RBD at Month 4-USA |  |  | 0.09 [0.03 to 2.28] | 0.42 [0.38 to 0.63] |  | 0.33 [0.25 to 0.41] | 0.15 [0.07 to 0.36]
  SARS-CoV-2 DB His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 DB His at Month 0-Peru |  | 1.64 [1.64 to 1.64] |  |  |  |  |
  SARS-CoV-2 DB His at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 18
  SARS-CoV-2 DB His at Month 0-Total | 1.55 [1 to 2.1] | 0.64 [0.35 to 1.14] | 0.06 [0.06 to 0.17] | 0.15 [0.06 to 1.1] | 0.18 [0.12 to 0.23] | 0.38 [0.22 to 0.83] | 0.62 [0.19 to 1.04]
  SARS-CoV-2 DB His at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 18
  SARS-CoV-2 DB His at Month 0-USA | 1.55 [1 to 2.1] | 0.35 [0.2 to 0.49] | 0.06 [0.06 to 0.17] | 0.15 [0.06 to 1.1] | 0.18 [0.12 to 0.23] | 0.38 [0.22 to 0.83] | 0.62 [0.19 to 1.04]
  SARS-CoV-2 DB His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 DB His at Month 2-Peru | 0.19 [0.12 to 0.49] | 0.08 [0.08 to 0.08] | 0.24 [0.14 to 0.6] | 0.09 [0.08 to 0.46] | 0.59 [0.26 to 2.59] | 9.18 [9.18 to 9.18] | 0.6 [0.46 to 1.51]
  SARS-CoV-2 DB His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 12
  SARS-CoV-2 DB His at Month 2-Total | 0.19 [0.13 to 0.64] | 0.07 [0.06 to 0.07] | 0.23 [0.07 to 0.71] | 0.35 [0.06 to 1.73] | 0.42 [0.29 to 2] | 6.59 [3.35 to 7.88] | 0.44 [0.19 to 1]
  SARS-CoV-2 DB His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 9
  SARS-CoV-2 DB His at Month 2-USA | 1.51 [1.51 to 1.51] | 0.06 [0.06 to 0.06] | 0.19 [0.08 to 0.78] | 0.62 [0.06 to 2.02] | 0.42 [0.42 to 0.42] | 3.35 [1.72 to 4.97] | 0.26 [0.18 to 0.96]
  SARS-CoV-2 DB His at Month 4-Peru: number analyzed (Participants) | 13 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 DB His at Month 4-Peru | 0.06 [0.06 to 0.29] | 0.06 [0.06 to 0.06] | 0.06 [0.06 to 0.08] | 0.66 [0.44 to 0.87] | 0.2 [0.08 to 1.51] | 1.64 [1.48 to 1.79] | 1.97 [1.27 to 3.36]
  SARS-CoV-2 DB His at Month 4-Total: number analyzed (Participants) | 13 | 1 | 8 | 6 | 6 | 4 | 11
  SARS-CoV-2 DB His at Month 4-Total | 0.06 [0.06 to 0.29] | 0.06 [0.06 to 0.06] | 0.1 [0.06 to 0.24] | 0.24 [0.1 to 0.5] | 0.2 [0.08 to 1.51] | 1.64 [1.08 to 2.16] | 1.27 [0.41 to 2.66]
  SARS-CoV-2 DB His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 4 | 0 | 2 | 6
  SARS-CoV-2 DB His at Month 4-USA |  |  | 0.25 [0.18 to 0.33] | 0.16 [0.06 to 0.34] |  | 1.57 [0.94 to 2.2] | 0.46 [0.2 to 1.35]
  SARS-CoV-2 Nucleoprotein His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 Nucleoprotein His at Month 0-Peru |  | 0.02 [0.02 to 0.02] |  |  |  |  |
  SARS-CoV-2 Nucleoprotein His at Month 0-Total: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 Nucleoprotein His at Month 0-Total | 1.58 [1.2 to 1.96] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.39] | 0.02 [0.02 to 0.02] | 0.3 [0.02 to 2.95] | 0.08 [0.02 to 0.64]
  SARS-CoV-2 Nucleoprotein His at Month 0-USA: number analyzed (Participants) | 2 | 1 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 Nucleoprotein His at Month 0-USA | 1.58 [1.2 to 1.96] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.39] | 0.02 [0.02 to 0.02] | 0.3 [0.02 to 2.95] | 0.08 [0.02 to 0.64]
  SARS-CoV-2 Nucleoprotein His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 Nucleoprotein His at Month 2-Peru | 0.02 [0.02 to 0.13] | 0.02 [0.02 to 0.02] | 0.08 [0.05 to 0.17] | 0.1 [0.06 to 0.21] | 0.27 [0.05 to 0.53] | 0.7 [0.7 to 0.7] | 0.06 [0.04 to 0.08]
  SARS-CoV-2 Nucleoprotein His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 Nucleoprotein His at Month 2-Total | 0.06 [0.02 to 0.19] | 0.02 [0.02 to 0.02] | 0.1 [0.02 to 0.52] | 0.02 [0.02 to 0.18] | 0.4 [0.08 to 0.59] | 0.7 [0.4 to 1.48] | 0.44 [0.03 to 0.72]
  SARS-CoV-2 Nucleoprotein His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 Nucleoprotein His at Month 2-USA | 2 [2 to 2] | 0.02 [0.02 to 0.02] | 0.25 [0.02 to 0.74] | 0.02 [0.02 to 0.12] | 0.96 [0.96 to 0.96] | 1.18 [0.64 to 1.72] | 0.51 [0.21 to 0.94]
  SARS-CoV-2 Nucleoprotein His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 Nucleoprotein His at Month 4-Peru | 0.02 [0.02 to 0.15] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.04] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.23] | 0.02 [0.02 to 0.02] | 0.1 [0.02 to 0.36]
  SARS-CoV-2 Nucleoprotein His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 Nucleoprotein His at Month 4-Total | 0.02 [0.02 to 0.15] | 0.02 [0.02 to 0.02] | 0.04 [0.02 to 0.12] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.23] | 0.57 [0.02 to 1.73] | 0.27 [0.02 to 0.5]
  SARS-CoV-2 Nucleoprotein His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 Nucleoprotein His at Month 4-USA |  |  | 0.13 [0.05 to 0.35] | 0.02 [0.02 to 0.02] |  | 2.35 [1.73 to 2.97] | 0.4 [0.09 to 1.16]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-Peru |  | 0.83 [0.83 to 0.83] |  |  |  |  |
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-Total: number analyzed (Participants) | 1 | 3 | 11 | 14 | 2 | 5 | 18
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-Total | 0.77 [0.77 to 0.77] | 0.03 [0.03 to 0.43] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.17] | 0.03 [0.03 to 0.03] | 0.08 [0.03 to 0.58] | 0.3 [0.05 to 0.5]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-USA: number analyzed (Participants) | 1 | 2 | 11 | 14 | 2 | 5 | 18
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 0-USA | 0.77 [0.77 to 0.77] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.17] | 0.03 [0.03 to 0.03] | 0.08 [0.03 to 0.58] | 0.3 [0.05 to 0.5]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-Peru: number analyzed (Participants) | 12 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-Peru | 0.03 [0.03 to 0.07] | 0.03 [0.03 to 0.03] | 0.17 [0.12 to 0.26] | 0.03 [0.03 to 0.37] | 0.24 [0.17 to 0.29] | 5.91 [5.91 to 5.91] | 0.18 [0.16 to 0.45]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-Total: number analyzed (Participants) | 13 | 2 | 17 | 14 | 7 | 3 | 14
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-Total | 0.03 [0.03 to 0.14] | 0.03 [0.03 to 0.03] | 0.1 [0.03 to 0.27] | 0.03 [0.03 to 0.24] | 0.19 [0.16 to 0.29] | 4.2 [2.12 to 5.05] | 0.26 [0.14 to 0.67]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-USA: number analyzed (Participants) | 1 | 1 | 10 | 11 | 1 | 2 | 11
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 2-USA | 0.36 [0.36 to 0.36] | 0.03 [0.03 to 0.03] | 0.05 [0.03 to 0.35] | 0.03 [0.03 to 0.24] | 0.16 [0.16 to 0.16] | 2.12 [1.07 to 3.16] | 0.33 [0.09 to 0.87]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 1 | 6 | 2 | 5
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-Peru | 0.03 [0.03 to 0.07] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.05] | 0.28 [0.28 to 0.28] | 0.08 [0.03 to 0.37] | 0.99 [0.79 to 1.18] | 0.6 [0.13 to 1.22]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 6 | 6 | 4 | 11
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-Total | 0.03 [0.03 to 0.07] | 0.03 [0.03 to 0.03] | 0.06 [0.03 to 0.12] | 0.03 [0.03 to 0.03] | 0.08 [0.03 to 0.37] | 0.99 [0.48 to 1.54] | 0.13 [0.08 to 0.91]
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 RBD-B.1.427/429-AB at Month 4-USA |  |  | 0.12 [0.08 to 0.19] | 0.03 [0.03 to 0.03] |  | 1.09 [0.61 to 1.57] | 0.08 [0.04 to 0.21]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-Peru |  | 0.81 [0.81 to 0.81] |  |  |  |  |
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-Total: number analyzed (Participants) | 1 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-Total | 0.23 [0.23 to 0.23] | 0.02 [0.02 to 0.42] | 0.02 [0.02 to 0.06] | 0.23 [0.02 to 0.68] | 0.84 [0.72 to 0.95] | 0.4 [0.15 to 0.92] | 0.44 [0.02 to 0.73]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-USA: number analyzed (Participants) | 1 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S Hexapro-293F-PPF at Month 0-USA | 0.23 [0.23 to 0.23] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.06] | 0.23 [0.02 to 0.68] | 0.84 [0.72 to 0.95] | 0.4 [0.15 to 0.92] | 0.44 [0.02 to 0.73]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-Peru | 0.1 [0.02 to 0.25] | 0.02 [0.02 to 0.02] | 0.15 [0.05 to 0.59] | 0.02 [0.02 to 0.02] | 0.72 [0.42 to 1.44] | 7.46 [7.46 to 7.46] | 0.4 [0.39 to 1.08]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-Total | 0.15 [0.03 to 0.47] | 0.02 [0.02 to 0.02] | 0.17 [0.04 to 0.64] | 0.02 [0.02 to 0.65] | 0.56 [0.34 to 1.25] | 0.5 [0.29 to 3.98] | 0.38 [0.02 to 0.87]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 S Hexapro-293F-PPF at Month 2-USA | 2.38 [2.38 to 2.38] | 0.02 [0.02 to 0.02] | 0.19 [0.05 to 0.85] | 0.02 [0.02 to 0.74] | 0.31 [0.31 to 0.31] | 0.29 [0.19 to 0.4] | 0.15 [0.02 to 0.73]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-Peru | 0.02 [0.02 to 0.29] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] | 0.12 [0.07 to 0.17] | 0.15 [0.04 to 0.71] | 1.57 [1.19 to 1.94] | 2.89 [1.25 to 3.01]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-Total | 0.02 [0.02 to 0.29] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.13] | 0.02 [0.02 to 0.09] | 0.15 [0.04 to 0.71] | 0.6 [0.35 to 1.19] | 0.46 [0.06 to 2.95]
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S Hexapro-293F-PPF at Month 4-USA |  |  | 0.16 [0.07 to 0.42] | 0.02 [0.02 to 0.02] |  | 0.31 [0.26 to 0.35] | 0.06 [0.02 to 0.37]
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-Peru |  | 1.15 [1.15 to 1.15] |  |  |  |  |
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-Total | 4.73 [2.48 to 6.98] | 0.02 [0.02 to 0.59] | 0.02 [0.02 to 0.14] | 0.42 [0.02 to 1.39] | 2.86 [1.63 to 4.08] | 0.53 [0.21 to 5.3] | 0.74 [0.1 to 1.93]
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-B.1.1.7-AB at Month 0-USA | 4.73 [2.48 to 6.98] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.14] | 0.42 [0.02 to 1.39] | 2.86 [1.63 to 4.08] | 0.53 [0.21 to 5.3] | 0.74 [0.1 to 1.93]
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-Peru | 0.19 [0.13 to 0.84] | 0.02 [0.02 to 0.02] | 0.24 [0.18 to 0.62] | 0.02 [0.02 to 0.02] | 1.27 [0.39 to 5.04] | 8.95 [8.95 to 8.95] | 1.01 [0.96 to 2.43]
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 13
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-Total | 0.3 [0.14 to 0.99] | 0.02 [0.02 to 0.02] | 0.25 [0.17 to 0.78] | 0.02 [0.02 to 1.31] | 0.51 [0.34 to 4.04] | 0.69 [0.39 to 4.82] | 0.75 [0.54 to 1.01]
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 10
  SARS-CoV-2 S-B.1.1.7-AB at Month 2-USA | 4.96 [4.96 to 4.96] | 0.02 [0.02 to 0.02] | 0.26 [0.1 to 0.72] | 0.25 [0.02 to 1.56] | 0.33 [0.33 to 0.33] | 0.39 [0.24 to 0.54] | 0.68 [0.48 to 0.92]
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-Peru | 0.09 [0.02 to 0.78] | 0.02 [0.02 to 0.02] | 0.06 [0.02 to 0.11] | 0.4 [0.21 to 0.59] | 0.41 [0.09 to 2.73] | 1.48 [1.21 to 1.76] | 4.35 [3.36 to 4.68]
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-Total | 0.09 [0.02 to 0.78] | 0.02 [0.02 to 0.02] | 0.12 [0.02 to 0.54] | 0.09 [0.02 to 0.43] | 0.41 [0.09 to 2.73] | 0.99 [0.77 to 1.29] | 0.74 [0.3 to 4.51]
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S-B.1.1.7-AB at Month 4-USA |  |  | 0.9 [0.15 to 2.04] | 0.09 [0.02 to 0.35] |  | 0.67 [0.48 to 0.86] | 0.3 [0.29 to 0.33]
  SARS-CoV-2 S-B.1.351-AB at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S-B.1.351-AB at Month 0-Peru |  | 1.47 [1.47 to 1.47] |  |  |  |  |
  SARS-CoV-2 S-B.1.351-AB at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-B.1.351-AB at Month 0-Total | 0.08 [0.04 to 0.12] | 0.01 [0.01 to 0.74] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.21] | 0.29 [0.28 to 0.29] | 0.08 [0.01 to 2] | 0.14 [0.01 to 0.49]
  SARS-CoV-2 S-B.1.351-AB at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-B.1.351-AB at Month 0-USA | 0.08 [0.04 to 0.12] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.21] | 0.29 [0.28 to 0.29] | 0.08 [0.01 to 2] | 0.14 [0.01 to 0.49]
  SARS-CoV-2 S-B.1.351-AB at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S-B.1.351-AB at Month 2-Peru | 0.01 [0.01 to 0.2] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.26] | 0.01 [0.01 to 0.01] | 0.62 [0.34 to 1.71] | 3.08 [3.08 to 3.08] | 0.12 [0.06 to 0.22]
  SARS-CoV-2 S-B.1.351-AB at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 S-B.1.351-AB at Month 2-Total | 0.03 [0.01 to 0.19] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.18] | 0.01 [0.01 to 0.09] | 0.53 [0.18 to 1.38] | 0.51 [0.26 to 1.8] | 0.13 [0.01 to 0.32]
  SARS-CoV-2 S-B.1.351-AB at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 S-B.1.351-AB at Month 2-USA | 0.18 [0.18 to 0.18] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.13] | 0.01 [0.01 to 0.32] | 0.09 [0.09 to 0.09] | 0.26 [0.14 to 0.39] | 0.14 [0.01 to 0.43]
  SARS-CoV-2 S-B.1.351-AB at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S-B.1.351-AB at Month 4-Peru | 0.01 [0.01 to 0.06] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.15 [0.08 to 0.22] | 0.2 [0.05 to 0.23] | 0.76 [0.51 to 1.02] | 0.18 [0.08 to 0.9]
  SARS-CoV-2 S-B.1.351-AB at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S-B.1.351-AB at Month 4-Total | 0.01 [0.01 to 0.06] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.15] | 0.2 [0.05 to 0.23] | 0.31 [0.24 to 0.59] | 0.09 [0.01 to 0.57]
  SARS-CoV-2 S-B.1.351-AB at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S-B.1.351-AB at Month 4-USA |  |  | 0.04 [0.01 to 0.22] | 0.01 [0.01 to 0.01] |  | 0.27 [0.23 to 0.32] | 0.05 [0.01 to 0.2]
  SARS-CoV-2 S-B.1.617-AB at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S-B.1.617-AB at Month 0-Peru |  | 1.34 [1.34 to 1.34] |  |  |  |  |
  SARS-CoV-2 S-B.1.617-AB at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 17
  SARS-CoV-2 S-B.1.617-AB at Month 0-Total | 0.34 [0.28 to 0.41] | 0.01 [0.01 to 0.67] | 0.01 [0.01 to 0.01] | 0.22 [0.01 to 0.38] | 0.27 [0.22 to 0.33] | 0.34 [0.14 to 2.73] | 0.32 [0.01 to 0.51]
  SARS-CoV-2 S-B.1.617-AB at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 17
  SARS-CoV-2 S-B.1.617-AB at Month 0-USA | 0.34 [0.28 to 0.41] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.22 [0.01 to 0.38] | 0.27 [0.22 to 0.33] | 0.34 [0.14 to 2.73] | 0.32 [0.01 to 0.51]
  SARS-CoV-2 S-B.1.617-AB at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S-B.1.617-AB at Month 2-Peru | 0.06 [0.01 to 0.16] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.35] | 0.01 [0.01 to 0.01] | 0.7 [0.35 to 1.98] | 4.17 [4.17 to 4.17] | 1.3 [0.74 to 1.71]
  SARS-CoV-2 S-B.1.617-AB at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 S-B.1.617-AB at Month 2-Total | 0.07 [0.01 to 0.29] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.26] | 0.01 [0.01 to 0.16] | 0.67 [0.19 to 1.57] | 0.42 [0.23 to 2.3] | 0.24 [0.05 to 1.11]
  SARS-CoV-2 S-B.1.617-AB at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 S-B.1.617-AB at Month 2-USA | 0.41 [0.41 to 0.41] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.25] | 0.01 [0.01 to 0.33] | 0.13 [0.13 to 0.13] | 0.23 [0.14 to 0.33] | 0.18 [0.01 to 0.44]
  SARS-CoV-2 S-B.1.617-AB at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S-B.1.617-AB at Month 4-Peru | 0.01 [0.01 to 0.11] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.07 [0.04 to 0.1] | 0.25 [0.06 to 0.36] | 0.65 [0.5 to 0.79] | 2.91 [0.12 to 3.31]
  SARS-CoV-2 S-B.1.617-AB at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S-B.1.617-AB at Month 4-Total | 0.01 [0.01 to 0.11] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.28] | 0.01 [0.01 to 0.01] | 0.25 [0.06 to 0.36] | 0.53 [0.27 to 0.76] | 0.24 [0.06 to 3.11]
  SARS-CoV-2 S-B.1.617-AB at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S-B.1.617-AB at Month 4-USA |  |  | 0.54 [0.01 to 1.39] | 0.01 [0.01 to 0.01] |  | 0.35 [0.18 to 0.53] | 0.12 [0.01 to 0.25]
  SARS-CoV-2 S-P.1-AB at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S-P.1-AB at Month 0-Peru |  | 1.43 [1.43 to 1.43] |  |  |  |  |
  SARS-CoV-2 S-P.1-AB at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-P.1-AB at Month 0-Total | 0.6 [0.51 to 0.69] | 0.04 [0.04 to 0.74] | 0.04 [0.04 to 0.15] | 0.45 [0.06 to 0.89] | 0.94 [0.66 to 1.22] | 0.91 [0.3 to 3.35] | 0.53 [0.06 to 1.6]
  SARS-CoV-2 S-P.1-AB at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 S-P.1-AB at Month 0-USA | 0.6 [0.51 to 0.69] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.15] | 0.45 [0.06 to 0.89] | 0.94 [0.66 to 1.22] | 0.91 [0.3 to 3.35] | 0.53 [0.06 to 1.6]
  SARS-CoV-2 S-P.1-AB at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S-P.1-AB at Month 2-Peru | 0.16 [0.12 to 0.53] | 0.1 [0.1 to 0.1] | 0.16 [0.07 to 0.33] | 0.04 [0.04 to 0.12] | 2.11 [0.58 to 4.02] | 3.57 [3.57 to 3.57] | 0.17 [0.16 to 0.78]
  SARS-CoV-2 S-P.1-AB at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 13
  SARS-CoV-2 S-P.1-AB at Month 2-Total | 0.21 [0.13 to 0.62] | 0.07 [0.05 to 0.08] | 0.18 [0.04 to 0.49] | 0.46 [0.04 to 1.64] | 0.62 [0.53 to 3.88] | 1.42 [0.79 to 2.49] | 0.37 [0.14 to 0.87]
  SARS-CoV-2 S-P.1-AB at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 10
  SARS-CoV-2 S-P.1-AB at Month 2-USA | 0.65 [0.65 to 0.65] | 0.04 [0.04 to 0.04] | 0.35 [0.04 to 0.51] | 1.4 [0.04 to 1.67] | 0.22 [0.22 to 0.22] | 0.79 [0.47 to 1.11] | 0.4 [0.11 to 0.8]
  SARS-CoV-2 S-P.1-AB at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S-P.1-AB at Month 4-Peru | 0.04 [0.04 to 0.4] | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.05] | 0.26 [0.15 to 0.37] | 0.89 [0.25 to 1.54] | 0.51 [0.44 to 0.59] | 0.19 [0.18 to 3.14]
  SARS-CoV-2 S-P.1-AB at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S-P.1-AB at Month 4-Total | 0.04 [0.04 to 0.4] | 0.04 [0.04 to 0.04] | 0.07 [0.04 to 0.43] | 0.41 [0.04 to 0.76] | 0.89 [0.25 to 1.54] | 0.62 [0.52 to 0.93] | 0.27 [0.17 to 1.88]
  SARS-CoV-2 S-P.1-AB at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S-P.1-AB at Month 4-USA |  |  | 0.57 [0.23 to 2.28] | 0.41 [0.04 to 1.05] |  | 1.15 [0.86 to 1.44] | 0.28 [0.1 to 0.54]
  SARS-CoV-2 S1 C His at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 S1 C His at Month 0-Peru |  | 1.08 [1.08 to 1.08] |  |  |  |  |
  SARS-CoV-2 S1 C His at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 13 | 2 | 5 | 19
  SARS-CoV-2 S1 C His at Month 0-Total | 0.61 [0.31 to 0.91] | 0.01 [0.01 to 0.55] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.18] | 0.09 [0.05 to 0.13] | 0.18 [0.01 to 0.71] | 0.32 [0.01 to 0.94]
  SARS-CoV-2 S1 C His at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 13 | 2 | 5 | 19
  SARS-CoV-2 S1 C His at Month 0-USA | 0.61 [0.31 to 0.91] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.18] | 0.09 [0.05 to 0.13] | 0.18 [0.01 to 0.71] | 0.32 [0.01 to 0.94]
  SARS-CoV-2 S1 C His at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 S1 C His at Month 2-Peru | 0.1 [0.01 to 0.21] | 0.01 [0.01 to 0.01] | 0.08 [0.01 to 0.29] | 0.01 [0.01 to 0.01] | 0.34 [0.07 to 2.42] | 7 [7 to 7] | 0.35 [0.22 to 1]
  SARS-CoV-2 S1 C His at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 S1 C His at Month 2-Total | 0.12 [0.01 to 0.26] | 0.01 [0.01 to 0.01] | 0.05 [0.01 to 0.34] | 0.01 [0.01 to 0.45] | 0.32 [0.12 to 1.76] | 3.66 [1.86 to 5.33] | 0.22 [0.01 to 1.02]
  SARS-CoV-2 S1 C His at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 S1 C His at Month 2-USA | 1.16 [1.16 to 1.16] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.36] | 0.01 [0.01 to 0.46] | 0.32 [0.32 to 0.32] | 1.86 [0.97 to 2.76] | 0.08 [0.01 to 1]
  SARS-CoV-2 S1 C His at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 S1 C His at Month 4-Peru | 0.01 [0.01 to 0.11] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.35 [0.18 to 0.52] | 0.01 [0.01 to 0.63] | 1.7 [1.29 to 2.1] | 1.28 [0.24 to 1.52]
  SARS-CoV-2 S1 C His at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 S1 C His at Month 4-Total | 0.01 [0.01 to 0.11] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.03] | 0.01 [0.01 to 0.22] | 0.01 [0.01 to 0.63] | 1.22 [0.7 to 1.79] | 0.27 [0.13 to 1.38]
  SARS-CoV-2 S1 C His at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 S1 C His at Month 4-USA |  |  | 0.04 [0.01 to 0.11] | 0.01 [0.01 to 0.01] |  | 0.84 [0.49 to 1.19] | 0.14 [0.01 to 0.42]
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-Peru |  | 3.34 [3.34 to 3.34] |  |  |  |  |
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-Total | 4.49 [3.7 to 5.28] | 2.39 [1.28 to 2.87] | 0.36 [0.21 to 0.54] | 2.16 [0.68 to 4.38] | 2.12 [2.11 to 2.13] | 1.91 [0.99 to 4.82] | 1.75 [0.71 to 4.4]
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2 spike (PreS Nexelis) at Month 0-USA | 4.49 [3.7 to 5.28] | 1.28 [0.73 to 1.84] | 0.36 [0.21 to 0.54] | 2.16 [0.68 to 4.38] | 2.12 [2.11 to 2.13] | 1.91 [0.99 to 4.82] | 1.75 [0.71 to 4.4]
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-Peru | 0.62 [0.32 to 1.3] | 0.18 [0.18 to 0.18] | 0.89 [0.29 to 1.18] | 0.39 [0.28 to 0.41] | 3.18 [0.99 to 6.52] | 13.71 [13.71 to 13.71] | 2.4 [1.82 to 3.39]
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-Total | 0.88 [0.35 to 1.69] | 0.18 [0.18 to 0.18] | 0.99 [0.28 to 1.26] | 1.53 [0.4 to 3.57] | 0.99 [0.96 to 6.14] | 7.53 [3.87 to 10.62] | 1.6 [1.24 to 2.25]
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2 spike (PreS Nexelis) at Month 2-USA | 3.85 [3.85 to 3.85] | 0.17 [0.17 to 0.17] | 1.09 [0.3 to 1.55] | 2.76 [1.21 to 4.82] | 0.57 [0.57 to 0.57] | 3.87 [2.05 to 5.7] | 1.54 [0.94 to 1.78]
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-Peru | 0.33 [0.17 to 1.3] | 0.17 [0.17 to 0.17] | 0.18 [0.17 to 0.19] | 1.08 [0.63 to 1.53] | 1.73 [0.59 to 4.58] | 2.29 [2.12 to 2.46] | 5.76 [3.42 to 8.19]
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-Total | 0.33 [0.17 to 1.3] | 0.17 [0.17 to 0.17] | 0.19 [0.17 to 0.61] | 1.94 [0.37 to 4.11] | 1.73 [0.59 to 4.58] | 2.72 [2.46 to 2.86] | 1.28 [0.81 to 6.97]
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2 spike (PreS Nexelis) at Month 4-USA |  |  | 0.76 [0.39 to 3.29] | 1.94 [0.56 to 6.25] |  | 2.92 [2.86 to 2.98] | 0.81 [0.6 to 1.17]
  SARS-CoV-2-NTD-AVI Biotin at Month 0-Peru: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SARS-CoV-2-NTD-AVI Biotin at Month 0-Peru |  | 0.1 [0.1 to 0.1] |  |  |  |  |
  SARS-CoV-2-NTD-AVI Biotin at Month 0-Total: number analyzed (Participants) | 2 | 3 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2-NTD-AVI Biotin at Month 0-Total | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.05] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.05] | 0.01 [0.01 to 0.01] | 0.22 [0.01 to 0.3] | 0.01 [0.01 to 0.32]
  SARS-CoV-2-NTD-AVI Biotin at Month 0-USA: number analyzed (Participants) | 2 | 2 | 11 | 15 | 2 | 5 | 19
  SARS-CoV-2-NTD-AVI Biotin at Month 0-USA | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.05] | 0.01 [0.01 to 0.01] | 0.22 [0.01 to 0.3] | 0.01 [0.01 to 0.32]
  SARS-CoV-2-NTD-AVI Biotin at Month 2-Peru: number analyzed (Participants) | 13 | 1 | 7 | 3 | 6 | 1 | 3
  SARS-CoV-2-NTD-AVI Biotin at Month 2-Peru | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.07] | 2.7 [2.7 to 2.7] | 0.01 [0.01 to 0.06]
  SARS-CoV-2-NTD-AVI Biotin at Month 2-Total: number analyzed (Participants) | 14 | 2 | 18 | 14 | 7 | 3 | 14
  SARS-CoV-2-NTD-AVI Biotin at Month 2-Total | 0.01 [0.01 to 0.05] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.11] | 0.19 [0.1 to 1.45] | 0.01 [0.01 to 0.14]
  SARS-CoV-2-NTD-AVI Biotin at Month 2-USA: number analyzed (Participants) | 1 | 1 | 11 | 11 | 1 | 2 | 11
  SARS-CoV-2-NTD-AVI Biotin at Month 2-USA | 0.06 [0.06 to 0.06] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.06] | 0.12 [0.12 to 0.12] | 0.1 [0.05 to 0.14] | 0.01 [0.01 to 0.17]
  SARS-CoV-2-NTD-AVI Biotin at Month 4-Peru: number analyzed (Participants) | 14 | 1 | 4 | 2 | 6 | 2 | 5
  SARS-CoV-2-NTD-AVI Biotin at Month 4-Peru | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.13 [0.07 to 0.19] | 0.01 [0.01 to 0.27]
  SARS-CoV-2-NTD-AVI Biotin at Month 4-Total: number analyzed (Participants) | 14 | 1 | 8 | 7 | 6 | 4 | 11
  SARS-CoV-2-NTD-AVI Biotin at Month 4-Total | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.11 [0.01 to 0.22] | 0.01 [0.01 to 0.08]
  SARS-CoV-2-NTD-AVI Biotin at Month 4-USA: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0 | 2 | 6
  SARS-CoV-2-NTD-AVI Biotin at Month 4-USA |  |  | 0.04 [0.01 to 0.07] | 0.01 [0.01 to 0.01] |  | 0.11 [0.06 to 0.16] | 0.01 [0.01 to 0.01]

64. Secondary Outcome: Detection of Viral RNA in Nasopharyngeal or Nasal Swab Samples Via RT-PCR
Description: This outcome measures the detection rate of viral RNA in nasopharyngeal or nasal swab samples collected at Visits 1, 2, 3, 4 using RT-PCR. Participation was optional, and not all participants provided samples. Results presented in this table include only participants from the Africa cohort (South Africa and other African countries), whose samples were tested using the RT-RNA Fisher TaqPath assay and Americas cohort (Peru and the United States), samples were tested using the RT-RNA Panther assay.
Time Frame: Measured at Months 0, Month 2, Month 4, Month 12
Population: Nasopharyngeal or nasal swab samples were collected at enrollment from 155 participants in the Americas cohort (Peru and USA) using the RT-RNA Panther assay, and from 320 participants in the Africa cohort (South Africa and other African countries) using the RT-RNA Fisher TaqPath assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 1C | Group 1D | Group 2A | Group 2B | Group 3
Number analyzed (Participants) | 81 | 36 | 122 | 49 | 83 | 43 | 61
Participants
  SARS-COV-2 IC at Month 0 Africa: number analyzed (Participants) | 69 | 12 | 98 | 23 | 66 | 19 | 22
  SARS-COV-2 IC at Month 0 Africa | 5 | 6 | 17 | 3 | 11 | 3 | 5
  SARS-COV-2 N-GENE at Month 0 Africa: number analyzed (Participants) | 69 | 12 | 98 | 23 | 66 | 19 | 22
  SARS-COV-2 N-GENE at Month 0 Africa | 5 | 6 | 17 | 3 | 11 | 3 | 5
  SARS-COV-2 ORF1ab at Month 0 Africa: number analyzed (Participants) | 69 | 12 | 98 | 23 | 66 | 19 | 22
  SARS-COV-2 ORF1ab at Month 0 Africa | 5 | 6 | 17 | 3 | 11 | 3 | 5
  SARS-COV-2 S-GENE at Month 0 Africa: number analyzed (Participants) | 69 | 12 | 98 | 23 | 66 | 19 | 22
  SARS-COV-2 S-GENE at Month 0 Africa | 5 | 6 | 17 | 3 | 11 | 3 | 5
  SARS-COV-2 IC at Month 2 Africa: number analyzed (Participants) | 0 | 2 | 1 | 3 | 1 | 2 | 1
  SARS-COV-2 IC at Month 2 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 N-GENE at Month 2 Africa: number analyzed (Participants) | 0 | 2 | 1 | 3 | 1 | 2 | 1
  SARS-COV-2 N-GENE at Month 2 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 ORF1ab at Month 2 Africa: number analyzed (Participants) | 0 | 2 | 1 | 3 | 1 | 2 | 1
  SARS-COV-2 ORF1ab at Month 2 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 S-GENE at Month 2 Africa: number analyzed (Participants) | 0 | 2 | 1 | 3 | 1 | 2 | 1
  SARS-COV-2 S-GENE at Month 2 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 IC at Month 4 Africa: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0
  SARS-COV-2 IC at Month 4 Africa | 0 | 0 | 1 | 0 | 0 | 0 | 0
  SARS-COV-2 N-GENE at Month 4 Africa: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0
  SARS-COV-2 N-GENE at Month 4 Africa | 0 | 0 | 1 | 0 | 0 | 0 | 0
  SARS-COV-2 ORF1ab at Month 4 Africa: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0
  SARS-COV-2 ORF1ab at Month 4 Africa | 0 | 0 | 1 | 0 | 0 | 0 | 0
  SARS-COV-2 S-GENE at Month 4 Africa: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0
  SARS-COV-2 S-GENE at Month 4 Africa | 0 | 0 | 1 | 0 | 0 | 0 | 0
  SARS-COV-2 IC at Month 12 Africa: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  SARS-COV-2 IC at Month 12 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 N-GENE at Month 12 Africa: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  SARS-COV-2 N-GENE at Month 12 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 ORF1ab at Month 12 Africa: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  SARS-COV-2 ORF1ab at Month 12 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SARS-COV-2 S-GENE at Month 12 Africa: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0
  SARS-COV-2 S-GENE at Month 12 Africa | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORF at Month 0 America: number analyzed (Participants) | 11 | 23 | 19 | 25 | 15 | 22 | 37
  ORF at Month 0 America | 0 | 1 | 0 | 0 | 0 | 0 | 1
  ORF at Month 2 America: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 0 | 1
  ORF at Month 2 America | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORF at Month 4 America: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ORF at Month 4 America | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ORF at Month 12 America: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ORF at Month 12 America | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected or assessed as part of the study
Description: Adverse Events were not collected or assessed as part of the study
Groups:
- Group 1: Persons not hospitalized for COVID-19, without clinical spectrum or outcomes specified in group 3
  * 1A: Persons with asymptomatic infection, ages 18 through 55, inclusive
  * 1B: Persons with asymptomatic infection, age > 55
  * 1C: Persons with symptomatic infection (ie, COVID-19) ages 18 through 55
  * 1D: Persons with symptomatic infection (ie, COVID-19), age > 55
  Sample collection: -Optional nasal specimen(s)
  -Blood collection
- Group 2: Persons previously hospitalized for COVID-19, without clinical spectrum or outcomes specified in group 3
  * 2A: Persons 18 through 55 years of age
  * 2B: Persons > 55 years of age
  Sample collection: -Optional nasal specimen(s)
  -Blood collection
- Group 3: Persons with specific clinical spectrums or outcomes, regardless of hospitalization history (eg, persons recovered after intubation, with prolonged viral shedding, with myocarditis/pericarditis, with rapid recovery from COVID-19, with a second positive SARS-CoV-2 RT-PCR test result after a negative result)
  Sample collection: -Optional nasal specimen(s)
  -Blood collection
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT04403880/Prot_SAP_ICF_000.pdf